

**Official Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

NCT Number: NCT00924703

Applicant/MAH: BioMarin Pharmaceutical Inc.

Version Date: 31 March 2017



#### CLINICAL STUDY PROTOCOL

Study Title: Long-term Extension of a Phase 2, Open-Label Dose-Finding Study

to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003

Investigational Product: rAvPAL-PEG
IND/EUDRACT Number: IND 076269
Indication: Phenylketonuria

**Sponsor:** BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

**Development Phase:** Phase 2

Sponsor's Responsible Medical Officer:

, MD , Clinical Affairs

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

**Duration:** Until product is commercially available or until study is terminated

**Dose:** 0.001 to 1.0 mg/kg per individual injection, with a maximum weekly

dose of 2.0 mg/kg

**Date of Original Protocol:** October 08, 2008

# Property of BioMarin CONFIDENTIAL

May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.

|--|

### 2 SYNOPSIS

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>rAvPAL-PEG | Volume:<br>Page:<br>Reference: | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

# PROTOCOL NUMBER: PAL-003

**STUDY SITES:** Approximately 8 centers in the United States

**PHASE OF DEVELOPMENT:** Phase 2

#### STUDY RATIONALE:

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve central nervous system developmental and functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding study (Study PAL-002). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

#### **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU who participated in Study PAL-002.
- To evaluate steady-state PK of rAvPAL-PEG in subjects with PKU.

#### STUDY DESIGN AND PLAN:

This is a long-term extension of a Phase 2, open-label, dose-finding study (Study PAL-002) in

| BIOMARIN <sup>®</sup> PAL-003 | OMARIN <sup>®</sup> |
|--------------------------------------------|---------------------|
|--------------------------------------------|---------------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>rAvPAL-PEG | Volume: Page: Reference: | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

approximately 35 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002.

Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

A Data Monitoring Committee will monitor the study.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 participants' rAvPAL-PEG dosing will continue in PAL-003 without interruption of weekly dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations below 480 µmol/L. Subjects will continue to receive injections in the clinic, administered by clinic staff, but may later be allowed to self-administer doses of study drug at home. Whether a subject may be allowed to self-administer study drug doses will be evaluated on an individual basis.

The dose may be modified at any time for safety.

Evaluations, observations, and procedures will be conducted at selected timepoints as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been controlled to within a target range (below 480  $\mu$ mol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses.

A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The drug becomes commercially available following the appropriate marketing approval.
- 4. The study is terminated.

| BIOMARIN | PAL-003 |
|----------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### Dose Adjustment Methodology:

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Depending upon the response to rAvPAL-PEG in PAL-002, a subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- The dose may be decreased as appropriate to achieve or maintain a favorable blood Phe concentration.
- When adjusting the dose, a dose may be used that is between the dose cohort levels that were defined in the previous study (PAL-002).
- The dose may be adjusted by increasing the frequency of injections per week, up to one dose per day, for a maximum total dose per week of 2 mg/kg.
- When a dose is adjusted (either by changing the dose level or by changing the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time.

Subjects must have blood Phe concentration tested 3 days after a dose adjustment. There must be a minimum of 2 weeks after each dose adjustment before any additional dose adjustments may be made, so that blood Phe concentrations can be assessed.

#### Stopping Criteria:

If an individual subject exhibits drug-related toxicity of CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level.

In addition, if 2 or more subjects at a dose level exhibit drug-related toxicity of CTCAE grade 3 or greater, further dosing of subjects at that dose level and any higher dose levels will be halted until a safety assessment is completed.

## **NUMBER OF SUBJECTS PLANNED:**

Approximately 35 subjects.

| PAL-003 |
|----------------------|
|----------------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>rAvPAL-PEG | Volume:<br>Page:<br>Reference: | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- Must have completed participation in PAL-002.
- Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- Willing and able to comply with all study procedures.
- Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- Maintained a stable diet.
- In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
- Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.

| BIOMARIN PAL-003 |
|-------------------------------|
|-------------------------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT: rAvPAL-PEG | Volume: Page: Reference: | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

- Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- Known hypersensitivity to rAvPAL-PEG or its excipients.
- Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- Creatinine > 1.5 times the upper limit of normal.

# INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

rAvPAL-PEG doses will be administered SC and the favorable dose (the dosage that provides control of blood Phe concentrations within the target range for a minimum of 2 weeks) will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses.

## **DURATION OF TREATMENT:**

Extension of multiple dosing will continue until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The drug becomes commercially available following the appropriate marketing approval.
- 4. The study is terminated.

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

| BIOMARIN | PAL-003 | |
|----------|---------|--------------|
| DICTIANT | PAL-003 | Page / 01 62 |

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### **CRITERIA FOR EVALUATION:**

# **Efficacy:**

Blood Phe concentrations will be measured.

#### Safety:

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs or laboratory test results.

#### **Pharmacokinetic:**

Plasma concentrations of rAvPAL-PEG will be measured when steady-state levels of Phe are attained.

### STATISTICAL METHODS:

#### Sample Size:

Subjects who participated in PAL-002 may be enrolled into this study. No formal sample size calculation was conducted.

#### Safety Analysis:

All subjects who receive any amount of study drug in this study will be included in the safety analyses.

Safety will be evaluated on the incidence of AEs, including serious AEs (SAEs), and clinically significant changes in vital signs and laboratory test results.

# **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any posttreatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled timepoint will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled timepoint will also be summarized.

#### **Pharmacokinetic Analysis:**

Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis.

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 480 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on

| BIOMARIN <sup>®</sup> PAL-003 |
|-------------------------------|
|-------------------------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |
| the same day each week for 3 consecutive weeks. | | |

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

# 2.1 Schedule of Events

**Table 2.1.1: Schedule of Events** 

| | Screening | | Treat | ment Period <sup>b,c</sup> | | Final F/U or<br>ETV |
|---|---|---|---|---|---|---|
| | | Week 1 | Weekly | Monthly (eg,<br>Wk 4, 8, etc, | Ortly (eg,<br>Wk 12, 24,<br>etc) | 4 weeks after<br>final dose |
| <b>Assessments and Events</b> | | D 1 | | | | |
| Informed consent | X | | | | | |
| Medical history and demographics | X | | | | | |
| Physical examination <sup>d</sup> | X | X | | | X | X |
| Vital signs | X | X | X | X | X | X |
| 12-lead ECG | X | | | | | X |
| Clinical laboratory tests <sup>e</sup> | X | | | X | X | X |
| Sedimentation rate | | X | | | X | X |
| Urine pregnancy test | X | X | | X | X | X |
| Injection-site inspectionf | | X<br>(postdose) | X | X | X | X |
| Adverse events <sup>g</sup> | Χ← | | | | | → X |
| Concomitant medications | X | X | X | X | X | X |
| Diet query | X | X | X | X | X | X |
| Serum rAvPAL-PEG antibodies | | X | | X | X | X |
| Predose blood Phe and plasma tyrosine <sup>h</sup> | X | X | X | X | X | X |
| Blood Phe (fingerstick) <sup>i</sup> | | | 3 days<br>postdos<br>e | | | |
| Predose PK sample <sup>j</sup> | | | | | | |
| Administer IP <sup>k</sup> | | X | X | X | X | |

AE, adverse event; D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> Screening assessments must be completed within 28 days from Day 1. These may be the same used for the Final Follow-up Visit of PAL-002, if they occur  $\leq$  28 days from Day 1.

<sup>&</sup>lt;sup>b</sup> Additional visits may occur if deemed necessary to monitor AEs or blood Phe, adjust dosing etc.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Complete physical examinations to include the evaluation of all major body systems, height (at Screening only), and weight.

<sup>&</sup>lt;sup>e</sup> Clinical laboratory tests to include hematology, chemistry, and urinalysis.

- f If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, e.g. right arm vs. left arm)
- <sup>g</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug to the final study visit.
- <sup>h</sup> Samples should be drawn in the morning, at least 2.5 hours after a meal. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.
- <sup>1</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.
- j. The PK blood samples will be collected after the subject has achieved and maintained target blood Phe concentration (below 480 μmol/L) for a minimum of 2 weeks. Once this target is achieved, predose PK samples will be collected on the same day each week for 3 consecutive weeks as specified in Section 9.7.3.
- <sup>k</sup> Dosing is up to 1.0 mg/kg per injection and up to one dose per day, for a total of up to 2.0 mg/kg/week.



PAL-003


# 3 TABLE OF CONTENTS

| 1 | TI | TLE PA | GE | 1 |
|---|---|---|---|---|
| 2 | SYN | NOPSIS. | | 2 |
| | 2.1 | Sched | ule of Events | 9 |
| 3 | TAE | BLE OF | CONTENTS | 11 |
| 4 | LIST | Γ OF AI | BBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 5 | ETH | IICS | | 19 |
| | 5.1 | Institu | tional Review Board or Ethics Committee | 19 |
| | 5.2 | Ethica | l Conduct of Study | 19 |
| | 5.3 | Subjec | ct Information and Informed Consent | 20 |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 21 |
| 7 | INT | RODUC | CTION | 22 |
| | 7.1 | Noncl | inical Studies | 22 |
| | 7.2 | Previo | ous Clinical Studies | 23 |
| | 7.3 | Study | Rationale | 23 |
| | 7.4 | Summ | nary of Overall Risks and Benefits | 24 |
| | | 7.4.1 | Toxicity Due to Exposure to PEG | 25 |
| | | 7.4.2 | Toxicity Due to Immunologic Sensitization | 25 |
| | | | 7.4.2.1 Management of Allergic Reactions | 26 |
| | | 7.4.3 | Effects of Low Blood Phe | 26 |
| 8 | STU | DY OB | JECTIVES | 27 |
| 9 | INV | ESTIGA | ATIONAL PLAN | 28 |
| | 9.1 | Overa | ll Study Design and Plan | 28 |
| | | 9.1.1 | Dose Adjustment Methodology | 29 |
| | | 9.1.2 | Stopping Criteria | 29 |
| | 9.2 | Discus | ssion of Study Design, Including Choice of Control Group | 30 |
| | 9.3 | Select | ion of Study Population | 30 |
| | | 9.3.1 | Inclusion Criteria | 30 |
| | | 9.3.2 | Exclusion Criteria | 31 |

| BIO | M | AF | 21 | N |
|-----|---|----|----|---|
|-----|---|----|----|---|

# PAL-003

# 

| | 9.3.3 Removal of Subjects from Treatment or Assessment | ent31 |
|-----|---------------------------------------------------------|-------|
| | 9.3.4 Subject Identification and Replacement of Subject | ts32 |
| 9.4 | Treatments | 33 |
| | 9.4.1 Treatments Administered | 33 |
| | 9.4.2 Identity of Investigational Product (IP) | 33 |
| | 9.4.2.1 Product Characteristics and Labeling | 33 |
| | 9.4.3 Storage | 33 |
| | 9.4.4 Directions for Administration | 33 |
| | 9.4.5 Method of Assigning Subjects to Treatment Group | ps34 |
| | 9.4.6 Selection of Doses Used in the Study | 34 |
| | 9.4.6.1 Selection of Timing of Dose for Each Subj | ect34 |
| | 9.4.7 Blinding | 34 |
| | 9.4.8 Prior and Concomitant Medications | 34 |
| | 9.4.9 Treatment Compliance | 35 |
| 9.5 | Investigational Product Accountability | 35 |
| | 9.5.1 Return and Disposition of Clinical Supplies | 35 |
| 9.6 | Dietary or Other Protocol Restrictions | 36 |
| 9.7 | Efficacy and Safety Variables | 36 |
| | 9.7.1 Efficacy and Safety Measurements Assessed | 36 |
| | 9.7.1.1 Demographic Data and Medical History | 36 |
| | 9.7.1.2 Physical Examination Findings | 36 |
| | 9.7.1.3 Vital Sign Measurements | 37 |
| | 9.7.1.4 Electrocardiography | 37 |
| | 9.7.2 Efficacy Variable | 37 |
| | 9.7.2.1 Blood Phenylalanine Concentrations | 37 |
| | 9.7.3 Pharmacokinetic Variables | 37 |
| | 9.7.4 Safety Variables | 37 |
| | 9.7.4.1 Pregnancy Testing | 37 |
| | 9.7.4.2 rAvPAL-PEG-specific Antibodies | |
| | 9.7.5 Clinical Laboratory Assessments | 38 |

| BION | 1AF | RIN |
|------|-----|-----|
|------|-----|-----|

# PAL-003


| 10 | REP | ORTING ADVERSE EVENTS | 40 |
|---|---|---|---|
| | 10.1 | Adverse Events | 40 |
| | 10.2 | Serious Adverse Events | 42 |
| | 10.3 | Pregnancy | 43 |
| | 10.4 | BioMarin Pharmacovigilance Contact Information | 43 |
| 11 | APP | ROPRIATENESS OF MEASUREMENTS | 44 |
| | 11.1 | Pharmacokinetics | 44 |
| 12 | STU | DY PROCEDURES | 45 |
| | 12.1 | Prestudy | 45 |
| | 12.2 | Screening Visit | 45 |
| | 12.3 | Treatment Period | 45 |
| | | 12.3.1 Day 1 (Week 1) | 46 |
| | | 12.3.2 Weekly Visits | 46 |
| | | 12.3.3 Monthly Visits (Week 4, 8, 16, etc) | 47 |
| | | 12.3.4 Quarterly Visits (Week 12, 24, 36, etc) | 47 |
| | 12.4 | Final Follow-up Visit (Day 113 [± 3 days]) /Early Termination Visit | |
| 13 | DAT | A QUALITY ASSURANCE | 49 |
| 14 | STA | TISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 50 |
| | 14.1 | Statistical and Analytical Plans | 50 |
| | 14.2 | Safety Analysis | 50 |
| | 14.3 | Pharmacokinetic Analysis | 50 |
| | 14.4 | Efficacy Analysis | 50 |
| | 14.5 | Determination of Sample Size | 51 |
| | | Handling of Missing Data | |
| | | Changes in the Conduct of the Study or Planned Analyses | |
| 15 | DAT | A MONITORING COMMITTEE (DMC) | 52 |
| | | IPENSATION, INSURANCE, AND INDEMNITY | |
| | | E REPORT FORMS AND SOURCE DOCUMENTS | |
| | | DY MONITORING AND AUDITING | |
| | | ENTION OF RECORDS | 57 |

| BIOMARIN | PAL-003 | |
|---|---|---|
| 20 USE OF INFORMATION | ON AND PUBLICATION | 58 |
| 21 REFERENCES | | 59 |
| 22 INVESTIGATOR RESI | PONSIBILITIES | 61 |
| 22.1 Conduct of Study | and Protection of Human Subjects | 61 |
| LIST OF TABLES | | |
| Table 2.1.1: Schedule of Ex | vents | 9 |
| Table 9.7.1.1: Summary of | Laboratory Assessments | 36 |
| Table 9.7.5.1: Clinical Labo | oratory Tests | 39 |



## 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase

AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

 $AUC_{0-7 \, days}$  area under the plasma concentration-time curve from time zero on Day 1 to

Day 8

BUN blood urea nitrogen

°C degree Celsius

C<sub>trough</sub> predose concentration of rAvPAL-PEG

CD Compact disk

CFR Code of Federal Regulations

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form

CTCAE Common Terminal Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure

DCF Data Clarification Form

DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

| BIOMARIN PAL-003 |
|--------------------------------|
|--------------------------------|

FDA Food and Drug Administration

f/u follow-up

g gram

GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure

IgG immunoglobulin G

IgM immunoglobulin M

ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IND Investigational New Drug

IP investigational product

IRB Institutional Review Board

IV intravenous

kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

NAb neutralizing antibodies

NCI National Cancer Institute

OTC over the counter

PAH phenylalanine hydroxylase

PAL phenylalanine ammonia lyase

| BIOMARIN | PAL-003 |
|----------|---------|
| BIOMARIN | PAL-003 |

PEG methoxypolyethylene glycol

Phe phenylalanine

PI Principal Investigator

PK pharmacokinetics

PKU phenylketonuria

rAvPAL-PEG phenylalanine ammonia lyase

RBC red blood cell

SAE serious adverse event

SAP Statistical Analysis Plan

SBP systolic blood pressure

SC subcutaneous

SD standard deviation

SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase

SGPT serum glutamic pyruvate transaminase

US United States

WBC white blood cell

| BIOMARIN | PAL-003 |
|----------|---------|

# Definition of Terms:

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.

| BIOMARIN PAL-003 |
|--------------------------------|
|--------------------------------|

### 5 ETHICS

### 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

# 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will

provide written, informed consent before any study-related tests or evaluations are performed.

# 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR §50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.

|--|

### 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Regulatory Affairs Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.

| PAL-003 |
|-----------------------|
|-----------------------|

### 7 INTRODUCTION

A comprehensive review of phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

# 7.1 Nonclinical Studies

The murine model of phenylketonuria (PKU) BTBRPah<sup>enu2</sup> (ENU<sup>2</sup>), a mouse line that is deficient in phenylalanine hydroxylase (PAH) activity (Shedlovsky, 1993, Genetics), was used for in vivo screening and pharmacodynamic studies. This mouse model exhibits characteristics similar to those seen in PKU patients, including hyperphenylalaninemia (baseline plasma phenylalanine [Phe] concentrations of 1000 to 2000 µM) and hypopigmentation. Weekly subcutaneous (SC) administration of 80 mg/kg of rAvPAL-PEG (approximately 4 IU/mouse) for greater than 3 months lowered blood Phe concentration from approximately 2000 μM to less than 200 μM. A similar profile of Phe reduction was also seen in ENU<sup>2</sup> mice administered wild-type AvPAL-PEG (4 IU/mouse) over 8 weeks. In all these studies, regardless of the molecule, an attenuated Phe-lowering response was usually seen between Weeks 2 and 7. However, plasma Phe concentrations became stabilized at concentrations below 200 µM from Week 7 onward. In addition to the reduction of plasma Phe, a dose-related darkening in coat color occurred, indicating the biosynthesis of melanin, which was previously inhibited when plasma Phe could not be metabolized and plasma Phe concentrations were high. When administration of AvPAL-PEG was stopped for 2 to 7 weeks and then reinitiated with weekly administrations, no attenuated response was observed and Phe concentrations remained low throughout the week.

The safety of rAvPAL-PEG was evaluated in safety pharmacology studies (respiratory, central nervous system [CNS] and cardiovascular [CV]) and toxicity with toxicokinetic studies (single and 28-day repeated dose) in rats and cynomolgus monkeys. Overall, in all toxicity studies no immune-related toxicities were seen either systemically or at the injection site. No specific methoxypolyethylene glycol (PEG)-related histological findings were observed during the 28-day repeated dose studies.

Findings in cynomolgus monkeys dosed with a single administration of 60 mg/kg rAvPAL-PEG included morbidity, decreased plasma Phe concentration, decreased protein synthesis, and gastrointestinal (GI) lesions. Plasma Phe concentrations were also reduced to below the level of detection in the lower dose groups, but without similar

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

toxicological consequence. Physiologically regulated Phe intake may have played a part in these morbidity results, although plasma Phe concentrations were low in all treated monkeys.

The main finding in the 28-day study was the possible drug-related observation of minimal to slight degeneration of blood vessels of predominantly medium-sized muscular arteries with a non-dose-dependent involvement of different organs observed in 1 male in the 0.1 mg/kg and 1 male and 1 female in the 1.0 mg/kg rAvPAL-PEG dose groups.

The half-life of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg, was 47, 33, and 44 hours, respectively, and exhibited modest area under the plasma concentration-time curve (AUC)-dose linearity. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the half-life was 65 hours at 4 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum plasma concentration, along with a long half-life, (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) AUC and the maximum plasma concentration (C<sub>max</sub>) are roughly linearly proportional.

### 7.2 Previous Clinical Studies

This study is an extension of the second human clinical study with rAvPAL-PEG (Study PAL-002). Study PAL-001, the first-in-human clinical study of rAvPAL-PEG, was designed as a Phase 1, open-label, single-dose, dose-escalation study in approximately 35 subjects, 16 to 50 years old, with PKU. The doses for this study are planned to be in the same range as those tested in PAL-001 and PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in those studies.

# 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH (Scriver CR, 2001, McGraw-Hill). Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver CR, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver CR, 2001, McGraw-Hill). The brains of untreated patients

| BIOMARIN | PAL-003 |
|----------|---------|

with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Leey, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan® is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve central nervous system developmental and functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding study (PAL-002). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

## 7.4 Summary of Overall Risks and Benefits

It is not expected that data from PAL-001 and PAL-002 will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

| BIOMARIN PAL-003 |
|--------------------------------|
|--------------------------------|

# 7.4.1 Toxicity Due to Exposure to PEG

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given up to 60 mg/kg of SC rAvPAL-PEG.

In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

# 7.4.2 Toxicity Due to Immunologic Sensitization

The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. In animal models, the immune response against the foreign protein PAL in rAvPAL-PEG has been mitigated by PEGylation. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylation does not eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing the immunogenicity of the molecule, it is reasonable to expect that some individuals may exhibit immune responses upon exposure to the drug. These immune responses may be clinically irrelevant, cause symptoms of various degrees, or lead to neutralization of biological activity. Subjects participating in clinical trials will be monitored closely with specific antibody titers, sedimentation rates, and complete blood counts (CBCs).

PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.) (Harris, 2003, Nat.Rev.Drug Discov.), and antibodies against PEG seem to form only under special circumstances (Harris, 2003, Nat.Rev.Drug.Discov.) (Richter, 1983, Int.Arch.Allergy Appl.Immunol.) and may be of no clinical relevance in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.).

Allergic reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 2 hours after injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of allergic reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection.

# 7.4.2.1 Management of Allergic Reactions

The following measures are recommended for the treatment of allergic symptoms:

- Clearing the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. Acetaminophen or ibuprofen (5-10 mg/kg) may also be administered. An allergy and/or immunology consultation should be sought if necessary.

#### 7.4.3 Effects of Low Blood Phe

Insufficient Phe intake or excessive rAvPAL-PEG exposure may cause blood Phe concentrations to be too low (eg,  $< 30 \mu mol/L$ ). Prolonged low blood Phe concentrations can result in a catabolic state associated with poor growth and altered body functions, including mental and physical alterations, loss of appetite, anemia, rashes, and diarrhea. To ensure safety during this study, subjects will be monitored closely with frequent blood Phe concentration determinations.

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

# 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU who participated in Study PAL-002.
- To evaluate steady-state PK of rAvPAL-PEG in subjects with PKU.

| BIOMARIN | PAL-003 |
|----------|---------|

### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of a Phase 2, open-label, dose-finding study (PAL-002) in approximately 35 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002.

Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

A Data Monitoring Committee will monitor the study.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 participants' rAvPAL-PEG dosing will continue in PAL-003 without interruption of weekly dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations below 480 µmol/L based upon recommendations by the German Working Group for Metabolic Diseases (Burgard, 1999, Eur J Pediatr). Subjects will continue to receive injections in the clinic, administered by clinic staff, but may later be allowed to self-administer doses of study drug at home. Whether a subject may be allowed to self-administer study drug doses will be evaluated on an individual basis. All of the following criteria must be met before a subject may self-administer doses of the study drug:

- The subject is willing and able to administer the study drug as directed.
- The sponsor agrees that self-administration is appropriate.
- The subject has achieved a favorable dose (ie, the dosage that provides control of blood Phe concentrations within the target range for a minimum of 2 weeks).
- The subject has received appropriate training, including administering doses under supervision, until the subject and clinic staff both agree such training is no longer necessary.

The dose may be modified at any time for safety.

Evaluations, observations, and procedures will be conducted at selected timepoints as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been

| BIOMARIN | PAL-003 |
|----------|---------|

controlled to within a target range (below 480 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses.

A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The drug becomes commercially available following the appropriate marketing approval.
- 4. The study is terminated.

# 9.1.1 Dose Adjustment Methodology

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Depending upon the response to rAvPAL-PEG in PAL-002, a subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- The dose may be decreased as appropriate to achieve or maintain a favorable blood Phe concentration.
- When adjusting the dose, a dose may be used that is between the dose cohort levels that were defined in the previous study (PAL-002).
- The dose may be adjusted by increasing the frequency of injections per week, up to one dose per day, for a maximum total dose of 2 mg/kg/week.
- When a dose is adjusted (either by changing the dose level or by changing the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time.

Subjects must have blood Phe concentration tested 3 days after a dose adjustment. There must be a minimum of 2 weeks after each dose adjustment before any additional dose adjustments may be made so that blood Phe concentrations can be assessed.

## 9.1.2 Stopping Criteria

If an individual subject exhibits drug-related toxicity of CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principle Investigator (PI) and the Study Medical Officer, and a decision

| BIOMARIN | PAL-003 |
|----------|---------|

will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level.

In addition, if 2 or more subjects at a dose level exhibit drug-related toxicity of CTCAE grade 3 or greater, further dosing of subjects at that dose level and any higher dose levels will be halted until a safety assessment is completed.

# 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

# 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- Must have completed participation in PAL-002.
- Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- Willing and able to comply with all study procedures.
- Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- Maintained a stable diet.
- In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

| BIOMARIN | PAL-003 |
|----------|---------|

#### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
- Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- Known hypersensitivity to rAvPAL-PEG or its excipients.
- Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- Creatinine > 1.5 times the upper limit of normal.

# 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study at any time without prejudice. The Investigator must withdraw from the study any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

| BIOMARIN | PAL-003 |
|----------|---------|

- Subject experiences a serious or intolerable AE.
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).

If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

# 9.3.4 Subject Identification and Replacement of Subjects

Each subject was assigned a unique subject identifier in either PAL-001 or PAL-002. Subjects will retain the same subject number used in PAL-002.

This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

| BIOMARIN | PAL-003 |
|----------|---------|

### 9.4 Treatments

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site with a supply of IP sufficient for the completion of the study.

## 9.4.2 Identity of Investigational Product (IP)

# 9.4.2.1 Product Characteristics and Labeling

The rAvPAL-PEG drug product for SC injection is formulated and supplied as a sterile aqueous (colorless to pale yellow) solution in clear, single-use, type-1 borosilicate glass vials. Each 3 mL vial contains  $1.5\pm0.2$  mL to deliver 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with  $1.5\pm0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Dilution instructions are provided in a separate instruction manual.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

Drug product packaging will be identified with the lot number and expiration date, and will be provided in a box labeled with the study number.

# 9.4.3 Storage

At the study site, all IP must be stored at  $5\pm3^{\circ}$ C ( $41\pm5^{\circ}$ F) under the conditions specified in the IB in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 2 mg/kg.

Dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous

measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

The injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

# 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in PAL-002.

# 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A favorable dose that produces a reduction in blood Phe concentration to below 480 µmol/L will be determined for each subject. Findings in cynomolgus monkeys dosed with a single administration of 60 mg/kg rAvPAL-PEG included severe morbidity, decreased plasma Phe concentration, decreased protein synthesis, and GI lesions. Plasma Phe concentrations were reduced to below the level of detection in the lower dose groups, without other findings. The doses for this study will be based upon the results of PAL-001 and PAL-002.

# 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered in the morning by clinic staff or by the subject, if appropriate.

### 9.4.7 Blinding

This is an open-label study.

# 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the medical monitor must be notified of the use of any

| BIOMARIN | PAL-003 |
|----------|---------|

contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in PAL-002) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

# 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

# 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

# 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.


## 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study except as necessary for safety.

# 9.7 Efficacy and Safety Variables

# 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis (Section 2.1) describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

Party Responsible for Section in Protocol for **Laboratory Assessment Performing Test Details** Central laboratory 9.7.5 Clinical laboratory tests rAvPAL-PEG-specific antibodies **BioMarin** 9.7.4.2 PK variables Central laboratory 9.7.3 Blood Phe concentrations Central laboratory 9.7.2.1

**Table 9.7.1.1: Summary of Laboratory Assessments** 

Phe, phenylalanine; PK, pharmacokinetic.

## 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

## 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of weight; general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Height will be measured at Screening only. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

| BIOMARIN PAL-003 |
|--------------------------------|
|--------------------------------|

## 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C).

# 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the final follow-up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

# 9.7.2 Efficacy Variable

## 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn in the morning, at least 2.5 hours after a meal, on the days and timepoints indicated in the Schedule of Events (Table 2.1.1).

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 480 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks.

BioMarin will perform the analysis.

## 9.7.4 Safety Variables

#### 9.7.4.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the timepoints specified in the Schedules of Events (Table 2.1.1). Female subjects with a positive pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test results.

Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

# 9.7.4.2 rAvPAL-PEG-specific Antibodies

Immunoglobulin G (IgG) and M (IgM) antibodies and neutralizing antibodies (NAb) to rAvPAL-PEG will be measured using validated immunogenicity assays at the timepoints indicated in the Schedules of Events (Table 2.1.1).

BioMarin will perform the analysis.

## 9.7.5 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.

Specific days for obtaining samples are provided in Table 2.1.1 and in Section 12. The scheduled clinical laboratory tests are listed in Table 9.7.5.1. A central laboratory will be used for analysis.

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

**Table 9.7.5.1: Clinical Laboratory Tests** 

| <b>Blood Chemistry</b> | Hematology | <b>Urine Tests</b> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if |
| Alkaline<br>Phosphatase | Hematocrit | Color | applicable |
| ALT (SGPT) | WBC count | рН | Pharmacokinetics |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Serum rAvPAL-PEG- |
| BUN | Differential cell count | Protein | specific antibodies |
| Creatinine | Sedimentation rate | Glucose | (IgG, IgM, and NAb) |
| GGT | | Bilirubin | |
| Total protein | | Nitrite | |
| Calcium | | Urobilinogen | |
| Sodium | | Hemoglobin | |
| Potassium | | | |
| Glucose | | | |
| Uric acid | | | |
| CO <sub>2</sub> | | | |
| Chloride | | | |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; CO<sub>2</sub>, carbon dioxide; GGT, gamma-glutamyltransferase; IgG, immunoglobulin G; IgM, immunoglobulin M; NAb, neutralizing antibodies; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.



#### 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

According to the ICH definition, an AE (or adverse experience) is "any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the IP."

An adverse drug reaction (ADR) is described by the ICH as "all noxious and unintended responses to a medicinal product related to any dose." This means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility, ie, the relationship cannot be ruled out.

An AE may include intercurrent illnesses or injuries that represent an exacerbation (increase in frequency, severity, or specificity) of pre-existing conditions (eg, worsening of asthma). Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The reporting period for non-serious AEs is the period from the first administration of study drug through the final F/U Visit or at the ETV. If a non-serious AE remains unresolved at the conclusion of the study, the PI and medical monitor will make a joint clinical assessment as to whether continued follow-up of the AE is warranted, and the results of this assessment must be documented. Resolution is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

The Investigator will assess AEs for severity, for relationship to IP, and as to whether the event meets one or more of the definitions of an SAE (refer to Section 10.2).

The Investigator will determine the severity of each AE and will record it on the source documents and AE CRF, using the categories defined below.

| Grade | Description |
|----------|-----------------------------------------|
| Mild | No limitation of usual activities |
| Moderate | Some limitation of usual activities |
| Severe | Inability to carry out usual activities |

| BIOMARIN | L-003 |
|----------|---------------------|
|----------|---------------------|

The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as "serious," which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the relationship of an AE to the IP and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably<br>Related | The administration of IP and the occurrence of the AE are reasonably related in time AND |
| | The AE is more likely explained by exposure to the IP than by other factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).

| BIOMARIN PAL-003 |
|--------------------------------|
|--------------------------------|

#### 10.2 Serious Adverse Events

A SAE is defined as any AE that:

- Results in death.
- Is life threatening, that is, places the subject at immediate risk of death from the event as it occurred. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires in-patient hospitalization or prolongation of an existing in-patient hospitalization. Admission of a subject to the hospital as an in-patient as a result of an AE, even if the subject is released on the same day, qualifies as hospitalization.
- Results in persistent or significant disability or incapacity. An event qualifies as
  resulting in a persistent or significant disability or incapacity if it involves a
  substantial disruption of the subject's ability to carry out usual life functions. This
  definition is not intended to include experiences of relatively minor or temporary
  medical significance.
- Is a congenital anomaly or birth defect, that is, an AE that occurs in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Is an important medical event that does not meet any of the above criteria, but may jeopardize the subject or require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such events are intensive treatment in the emergency room, allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

More than one of the above criteria may apply to any specific event.

The reporting period for SAEs begins earlier than non-serious AEs and is the period from the time of signing of the ICF through 4 weeks after the last dose or at the ETV. SAEs reported to the Investigator outside of this reporting period will be reported to BioMarin if, in good medical judgment, the event has any bearing on the study data. SAEs must be followed by the Investigator until resolution, even if this extends beyond the study-reporting period. Resolution of an SAE is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

Any SAE, whether or not considered related to study drug, will be reported immediately (within 24 hours) to BioMarin Pharmacovigilance by fax using the study-specific SAE Report Form. In addition to the outcome of the SAE, any medication or other therapeutic measures used to treat the event will be recorded on the appropriate CRF page(s). Investigators should not wait to collect additional information that fully documents the event before notifying BioMarin Pharmacovigilance of an SAE. BioMarin may be required to



report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit additional information requested by BioMarin as soon as it becomes available.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

#### 10.3 Pregnancy

Pregnancy in a subject or partner should be reported immediately (within 24 hours) to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up Form in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

## 10.4 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the medical monitor any AEs for which the issue of seriousness is unclear or questioned. Contact information for the medical monitor is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone: Fax:

E-mail:

| BIOMARIN PAL-003 |
|--------------------------------|
|--------------------------------|

# 11 APPROPRIATENESS OF MEASUREMENTS

# 11.1 Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

#### 12 STUDY PROCEDURES

# 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

## 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history and demographics
- Physical examination and height
- Vital signs
- 12-lead ECG
- Clinical laboratory tests (including hematology, chemistry, and urinalysis)
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration

For subjects who participated in PAL-002, these assessments may be the same used for the Final Follow-up Visit of PAL-002, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done on the third day following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

| BIOMARIN PAL-003 | OMARIN |
|--------------------------------|--------|
|--------------------------------|--------|

## 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (postdose)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies
- Administer study drug (study drug may be administered on additional days during the week [up to 1 dose per day] as determined by the Investigator, in agreement with the Study Medical Officer)

## 12.3.2 Weekly Visits

The following study activities will be performed at the weekly visits beginning with Week 2:

- Vital signs
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasm tyrosine concentration
- Administer study drug (study drug may be administered on additional days during the week [up to 1 dose per day] as determined by the Investigator, in agreement with the Study Medical Officer)

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

| BIOMARIN | PAL-003 |
|----------|---------|

## 12.3.3 Monthly Visits (Week 4, 8, 16, etc)

The following study activities will be performed at the monthly visits beginning with Week 4:

- Vital signs
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies
- Administer study drug (study drug may be administered on additional days during the week [up to 1 dose per day] as determined by the Investigator, in agreement with the Study Medical Officer)

## 12.3.4 Quarterly Visits (Week 12, 24, 36, etc)

Quarterly visits consist of all monthly activities and include additional activities. The following study activities will be performed at the quarterly visits beginning with Week 12:

- Physical examination
- Vital signs
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration

| BIOMARIN | PAL-003 |
|----------|---------|

- Serum rAvPAL-PEG antibodies
- Administer study drug (study drug may be administered on additional days during the week [up to 1 dose per day] as determined by the Investigator, in agreement with the Study Medical Officer)

## 12.4 Final Follow-up Visit (Day 113 [± 3 days]) /Early Termination Visit

The final follow-up (F/U) Visit or Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the F/U Visit or ETV:

- Physical examination and weight
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies

| BIOMARIN | PAL-003 |
|----------|---------|

# 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

# 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

## 14.2 Safety Analysis

All subjects who receive any amount of study drug will be included in the safety analyses.

Safety will be evaluated on the incidence of AEs and clinically significant changes in vital signs and laboratory test results.

The verbatim terms reported on CRFs to identify AEs will be coded using MedDRA. Treatment-emergent AEs will be summarized for each treatment group by system organ class, preferred term, relationship to study drug, and severity. Changes from baseline in vital signs and laboratory test results will be summarized with descriptive statistics by dose group.

## 14.3 Pharmacokinetic Analysis

Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis.

Steady-state PK of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 480  $\mu$ mol/L) for a minimum of 2 weeks and no further dose modification is planned.

#### 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any posttreatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled timepoint will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled timepoint will also be summarized.

#### 14.5 Determination of Sample Size

Subjects who participated in PAL-002 may be enrolled into this study. No formal sample size calculation was conducted.

## 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.

# 14.7 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.

| BIOMARIN | PAL-003 |
|----------|---------|

## 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act in an advisory capacity to BioMarin to monitor subject safety and the efficacy of rAvPAL-PEG in subjects who participate in the study. Meetings of the DMC can be convened at any time at the discretion of the DMC Chair or the Study Medical Officer. The Chair will be notified by the Study Medical Officer of all SAEs and will receive summaries of other safety data as available. The DMC will review the study data as soon as it is available during the study and offer advice on whether or not to close the study on the basis of toxicity. Details regarding the DMC membership and safety data to be reviewed by members will be provided in a charter.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping rules as defined in study protocol.

| BIOMARIN | PAL-003 |
|----------|---------|

## 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries. The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment. If the subject has followed the Investigator's instructions, BioMarin will pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures, if these costs are not covered by health insurance or another third party that usually pays these costs. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.

| BIOMARIN | PAL-003 |
|----------|---------|

#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent. If an Investigator or institution refuses to allow access to subject records because of confidentiality, arrangements must be made to allow an "interview" style of data verification.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.

| BIOMARIN | PAL-003 |
|----------|---------|

#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (eg, subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.

|--|

## 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.

| PAL-003 |
|-----------------------|
|-----------------------|

#### 21 REFERENCES

Armstrong, Hempel, Koling, Chan, Fisher, Meiselman, Garratty. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007.

Burgard, Bremer, Bührdel, Clemens, Mönch, Przyrembel, Trefz, Ullrich. Rationale for the German recommendations for phenylalanine level control in phenylketonuria 1997. Eur J Pediatr 158, 46-54. 1999.

Butterworth. Effects of hyperammonaemia on brain function. J Inherit Metab Dis 21 Suppl 1, 6-20, 1998.

Chen, Scott. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001.

Davis, Abuchowski, Park, Davis. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981.

Fisch. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000.

Gamez, Wang, Sarkissian, Wendt, Fitzpatrick, Lemontt, Scriver, Stevens. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007.

Ganson, Kelly, Scarlett, Sundy, Hershfield. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006.

Guttler, Azen, Guldberg, Romstad, Hanley, Levy, Matalon, Rouse, Trefz, de la, Koch. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003.

Harris, Chess. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003.

Huttenlocher. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000.

Kaufman. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989.

Koch, Hanley, Levy, Matalon, Matalon, Rouse, Trefz, Guttler, Azen, Platt, Waisbren, Widaman, Ning, Friedman, de la. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003.

Lee, Lilburn, Baudin. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003.

Levy. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003.

Matalon, Surendran, Matalon, Tyring, Quast, Jinga, Ezell, Szucs. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003.

Richter, Akerblom. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983.

Richter, Akerblom. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984.

Rouse, Azen. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004.

Scott, Murad, Koumpouras, Talbot, Eaton. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997.

Scriver CR, Kaufman S. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-709.

Shedlovsky, McDonald, Symula, Dove. Mouse models of human phenylketonuria. Genetics 134[4], 1205-1210. 1993.

Walter, White, Hall, MacDonald, Rylance, Boneh, Francis, Shortland, Schmidt, Vail. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002.

Webster, Didier, Harris, Siegel, Stadler, Tilbury, Smith. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007.

#### 22 INVESTIGATOR RESPONSIBILITIES

# 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.

| BIOMARIN | PAL-003 |
|----------|---------|
| 1 | |

#### 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

**Protocol Number: PAL-003** 

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

| Investigator | Signature | Date |
|---------------|-----------|------|
| Printed name: | | |

## Accepted for the Sponsor:

On behalf of BioMarin, I confirm that BioMarin, as a sponsor will comply with all obligations as detailed in all applicable regulations and guidelines. I will ensure that the PI is informed of all relevant information that becomes available during the conduct of this study.

| | 10/16/2008 |
|-----------------|------------|
| Medical Monitor | Date |
| Printed name: | |




# CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Study Title: Long-term Extension of a Phase 2, Open-Label Dose-Finding

> Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with

**PKU** 

**Protocol Number: PAL-003** 

**Investigational Product:** rAvPAL-PEG

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria

BioMarin Pharmaceutical Inc. Sponsor:

> 105 Digital Drive Novato, CA 94949

**Development Phase:** Phase 2

Sponsor's Responsible

, MD , Clinical Affairs Medical Officer:

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

**Duration:** Until product is commercially available or until study is

terminated

0.001 to 1.0 mg/kg per individual injection, with a maximum Dose:

weekly dose of 2.0 mg/kg

**Date of Original Protocol:** October 08, 2008

Date of Amendment 1: February 09, 2009

Property of BioMarin

CONFIDENTIAL

May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.




#### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Amendment: 1

Date: February 09, 2009

#### RATIONALE AND SUMMARY OF CHANGES

The protocol has been amended as follows:

- Prohibited the use of polyethylene glycol (PEG)-containing injectable medications, because of reported unexpected adverse events (AEs) after intramuscular Depo-Provera<sup>®</sup> injection in 2 subjects.
- Excluded subjects taking or planning to take PEG-containing injectable medications.
- Added a list of PEG-containing injectable medications as an appendix to the protocol.
   This list is subject to change.
  - Provided details regarding the 2 subjects who experienced a study drug injection-site reaction and developed unexpected hypersensitivity AEs after a Depo-Provera injection (15 and 40 days, respectively) after the rAvPAL-PEG injection.
  - 3. Added the provision that subjects who experience an allergic reaction may be asked to see an allergist/immunologist and/or provide additional blood samples for antibody testing.
  - 4. Clarified that subjects may require more than 1 injection per dose, depending upon site policy.
    - Added a table as an example.
  - 5.
  - Added that at least one interim analysis may be performed by the Sponsor.
  - In interactive voice response system (IVRS) will be track subjects' assigned dose and study drug inventory.
  - 8. Provided clarifying language to allow subjects to complete PAL-002 study and enroll into PAL-003 without study drug interruption.
  - Specified there will be replacement of subjects in this study if any single cohort (identified during PAL-002) drops to less than 3 subjects after the initial enrollment of 35.



- 10. Made revisions to correct spelling, spacing, or punctuation, and/or made minor editorial revisions to improve clarity and consistency.
- 11. PAL-001 and/or PAL-002 data may become available during this study and indicate the need for pharmacokinetic measurement of study drug accumulation (in addition to the current plan for analysis of study drug exposure). If this is the case, the PAL-003 protocol will be amended to require additional blood draws for PK analysis.

| BIOMARIN |
|----------|
|----------|


# PROTOCOL AMENDMENT TEXT REVISIONS

The following table summarizes the revisions made to the protocol and relates the changes to the appropriate rationale. Text that has been added or inserted is indicated by <u>underlined</u> font, and deleted text is indicated by <u>strikethrough</u> font.

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| Section 2 Synopsis (Study Rationale) | STUDY RATIONALE: The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve central nervous system developmental and functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study will build upon the results of the first single-dose pharmacokinetics (PK) study (Study PAL-001) and evaluate whether weekly injections of rAvPAL-PEG can reduce blood Phe concentrations in PKU subjects and whether repeated administration is safe. | | 10 |
| Section 2 Synopsis<br>(Diagnosis and All<br>Criteria for Inclusion<br>and Exclusion) | <ul> <li>Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:</li> <li>Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.</li> <li>Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.</li> </ul> | | 1 |

 February 09, 2009




| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation. | | |
| | <ul> <li>A prior reaction that included systemic symptoms (eg, generalized hives,<br/>respiratory or gastrointestinal problems, hypotension, angioedema,<br/>anaphylaxis) to rAvPAL-PEG or a PEG-containing product.</li> </ul> | | |
| | <ul> <li>Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).</li> <li>Any condition that in the view of the PL places the subject at high risk of</li> </ul> | | |
| | <ul> <li>Any condition that, in the view of the PI, places the subject at high risk of<br/>poor treatment compliance or of not completing the study.</li> </ul> | | |
| Table 2.1.1 Schedule of Events (footnote a) | <sup>a</sup> It is preferable to perform PAL-003 Screening assessments the same day as PAL-002 Final Follow-up Visit so there is no interruption of study drug. If performed on the same day, PAL-002 Final Follow-up Visit data may be used. If not, PAL-003 Day 1 must occur ≤ 28 days after PAL-003 Screening. | | 8 |

 February 09, 2009




| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Section 4 List of<br>Abbreviations and<br>Definitions of Terms | IM intramuscular | Added new term | 10 |
| Section 4 List of<br>Abbreviations and<br>Definitions of Terms | IVRS interactive voice response system | Added new term | 7 |
| Section 4 List of<br>Abbreviations and<br>Definitions of Terms | PEG methoxypolyethylene glycol | | 10 |
| Section 7.1<br>Nonclinical Studies | When administration of AvPAL-PEG was stopped for 2 to 7 weeks and then reinitiated with weekly administrations, no attenuated response was observed and Phe concentrations remained low and stable until the next administration throughout the week. | Paragraph 1 | 10 |
| Section 7.1<br>Nonclinical Studies | No specific methoxypolyethylene glycol (PEG)-related histological findings were observed during the 28-day repeated dose studies. | Paragraph 2 | 10 |
| Section 7.1<br>Nonclinical Studies | Findings in cynomolgus monkeys dosed with a single administration of 60 mg/kg rAvPAL-PEG included morbidity, reduced food consumption, dehydration, body weight loss, hypoactivity, hypothermia, decreased plasma Phe concentration, decreased protein synthesis, and gastrointestinal (GI) lesions. Plasma Phe concentrations were also reduced to below the level of detection in the lower 4 and 12 mg/kg dose groups, but without similar toxicological consequence, implying that the physiological regulation of Phe levels may be an important factor for influencing morbidity. Physiologically regulated Phe intake may have played a | Paragraphs 4 and 5 | 10 |





| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | part in these morbidity results, although plasma Phe concentrations were low in all treated monkeys. | | |
| | The main finding in the 28-day study was the possible drug-related observation of minimal to slight degeneration of blood vessels of predominantly medium-sized muscular arteries with a non-dose-dependent involvement of different organs observed in 1 male in the 0.1 mg/kg and 1 male and 1 female in the 1.0 mg/kg rAvPAL-PEG dose groups. No degeneration of the arteries was observed in animals administered 0 and 0.01 mg/kg rAvPAL-PEG. | | |
| Section 7.3 Study<br>Rationale | The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood Phe concentrations and improve CNS developmental and functional outcomes. rAvPAL-PEG is a potential substitute for the PAH enzyme. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study will build upon the results of PAL-001 and evaluate whether weekly injections of rAvPAL-PEG can reduce blood Phe concentrations in PKU subjects and whether repeated administration is safe. | | 10 |

 February 09, 2009




| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Section No./Title Section 7.4.2 Toxicity Due to an Immunologic Reaction | PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.) (Harris, 2003, Nat.Rev.Drug Discov.), and however, antibodies against PEG seem to form only under special circumstances may form when PEG is bound to compounds. (Harris, 2003, Nat.Rev.Drug.Discov.) (Richter, 1983, Int.Arch.Allergy Appl.Immunol.) and may be of no In some instances, development of such antibodies did not result in any significant clinical relevance effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.). Two subjects enrolled in PAL-001 who had received one dose of rAvPAL-PEG experienced hypersensitivity reactions to intramuscular (IM) Depo-Provera, a contraceptive containing PEG 3350. Both subjects had previously received multiple IM Depo-Provera injections without complications. The first subject, a year old developed bruising at the injection site on Day 1 that resolved on Day 15. | Comments | Change No. 2, 3, 10 |
| | 10 minutes after receiving IM Depo-Provera and 40 days after rAvPAL-PEG injection. was treated in the emergency room with . The events resolved the same day, and the subject had no further complications. The subject had no prior history of any reactions to Depo-Provera. Subsequently, while under the care of an allergist/immunologist, the subject had a mild reaction to a concentrated intradermal (1:10) exposure of Depo-Provera. was later given a full dose of IM Depo-Provera without problems. | | |


**B**OMARIN

**PAL-003** 


| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | The second subject, an year old , had a slightly raised, erythematic rash | | |
| | below the site of rAvPAL-PEG injection on Day 11 that resolved without treatment | | |
| | on Day 15. developed generalized hives on arms and legs and mild | | |
| | difficulty breathing 20 minutes after receiving IM Depo-Provera (and third dose | | |
| | of Gardasil) given 15 days after rAvPAL-PEG injection. symptoms | | |
| | subsided after received given by mother. did not visit the | | |
| | emergency room. The subject had no prior history of any reactions to Depo-Provera | | |
| | or Gardasil (Gardasil dose not contain PEG). was subsequently seen by an | | |
| | allergist/immunologist, and the results are pending. | | |
| | Because Depo-Provera contains PEG 3350 as an excipient, it is possible that the administration of rAvPAL-PEG caused anti-PEG antibody formation that led to a cross-reaction with Depo-Provera in these subjects. Therefore, it is possible that prior exposure to rAvPAL-PEG might sensitize subjects to other PEG-containing injectable drugs. Alternatively, the presence of Depo-Provera could have led to antibody formation and cross-reaction with rAvPAL-PEG, leading to rAvPAL-PEG injection-site reactions. Since it is currently unknown whether Depo-Provera has a sensitizing effect to PEG and the exact basis for these reported events is not known, the use of PEG-containing injectable drugs prior to and during the study is prohibited as a precautionary measure (refer to the addendum and Sections 9.3.2 and 9.4.8). | | |
| | In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for antibody testing. This additional testing may occur up to 6 months following the final study visit. | | |



| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Section 9.1.1 | 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEG | Added new | 5 |
| Management of Local | 9.1.1.1 Subjects Who Have Experienced Hypersensitivity Reactions to | section | |
| and Systemic | rAvPAL-PEG or a PEG-containing Product | | |
| Reactions to rAvPAL- | Subjects who had a previous reaction to rAvPAL-PEG or a PEG-containing | | |
| PEG | product that warranted early termination from PAL-001 or PAL-002 are excluded | | |
| | from this study. However, subjects may develop such reactions after enrollment in | | |
| | PAL-003. Management of such reactions are described below. Refer to | | |
| | Figure 9.1.1.1.2.1: for a flowchart for managing these subjects. | | |
| | 9.1.1.2.1 Subjects with Local Reactions | | |
| | After enrollment in PAL-003, subjects who have a local reaction to rAvPAL-PEG | | |
| | or a PEG-containing product will be premedicated with acetaminophpen and | | |
| | antihistamines and/or oral steroids, 1 hour prior to study drug dosing. | | |
| | Recommended premedications are acetaminophen and antihistamine (Claritin is | | |
| | preferred). The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg | | |
| | Claritin or 25 to 50 mg oral Benadryl; an example for steroids would be 70 mg oral | | |
| | prednisone). Because Benadryl can cause drowsiness, it should be administered only if the subject is accompanied by a designated driver. | | |
| | 9.1.1.2.2 Subjects with Systemic Reactions | | |
| | After enrollment in PAL-003, subjects who have a systemic reaction that includes | | |
| | noncutaneous systemic symptoms, such as respiratory problems, hypotension, or | | |
| | angioedema, to rAvPAL-PEG or a PEG-containing product will be evaluated with a skin prick test. If the test is positive, the subject will be excluded from the study. | | |
| | Subjects with prior systemic reactions that included only skin manifestations to rAvPAL-PEG or a PEG-containing product after PAL-003 enrollment will be | | |
| | premedicated with acetaminophen and antihistamines and/or oral steroids (one hour | | |
| | prior to study drug dosing) and will continue to receive rAvPAL-PEG. | | |
| | prior to study drug dosing, and will continue to receive IAVI AL-1 LG. | | |




| Section No./Title | Reactions to skin prick testing or rAvPAL-PEG administered SC are defined as follows: Local reaction: 1 affected location, ie, hives, wheals, or swelling or an area of erythema or redness at or near the site of injection. Systemic reaction: more than 1 affected location, ie, cutaneous reaction in more than 1 area, and/or any other generalized symptoms, such as hypotension, angioedema or anaphylaxis or the involvement of other organ systems (eg, respiratory, cardiovascular, gastrointestinal). | Comments | Relates to<br>Change No. |
|---|---|---|---|
| Section 9.1.1 Management of Local and Systemic Reactions to rAvPAL- PEG | Figure 9.1.1.2.1 Management of Local and System Reactions to rAvPAL-PEG | Added new figure | 5 |
| Section 9.3.2<br>Exclusion Criteria | <ul> <li>Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study: <ul> <li>Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.</li> </ul> </li> <li>Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.</li> </ul> | | 1 |





| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | <ul> <li>A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product.</li> </ul> | | |
| | • Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug. | | |
| | <ul> <li>Pregnant or breastfeeding at Screening or planning to become pregnant (self<br/>or partner) or to breastfeed at any time during the study.</li> </ul> | | |
| | <ul> <li>Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).</li> </ul> | | |
| | <ul> <li>Any condition that, in the view of the PI, places the subject at high risk of<br/>poor treatment compliance or of not completing the study.</li> </ul> | | |
| Section 9.3.4 Subject<br>Identification and<br>Replacement of<br>Subjects | After enrollment of 35 subjects, if any single cohort (identified during PAL-002) has less than 3 subjects due to early terminations, those subjects will be replaced. Replacement subjects will enter the study at the same dose cohort level as the subject they are replacing. | | 9 |

 February 09, 2009




| Section No./Title | Revision | | | | Comments | Relates to Change No. |
|---|---|---|---|---|---|---|
| Section 9.4.4 Directions for Administration | Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). The number of injections required for an individual weighing 80 kg (about 176 pounds) is provided in Table 9.4.4.1 as an example. Note this table is for example purposes only. Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Table 9.4.4.1: Number of Injections Required For an Individual Weighing 80 kg | | | | | 4 |
| | Dose Group (mg/kg) 0.001 0.003 0.01 0.03 0.1 0.3 1.0 | Weight (kg) 80 8 | Volume of Study Drug (mL) <sup>a</sup> 0.8 0.6 0.8 0.2 0.8 2.4 8.0 | $ \frac{\text{No. of}}{\text{Injections}^{b}} $ $ \frac{1}{1} $ $ \frac{1}{2} $ $ \frac{1}{4} $ | | |
| | as specified in the PAI starting volume attains | at a concentration of 2-003 Pharmacy March following dilution er dose is dependent | 10 mg/mL and is then diluted by nual. Volume to be injected is call. upon site policy for SC injection | / differential amounts<br>lculated based on a | | |





| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Section 9.4.5 Method of Assigning Subjects to Treatment Groups | An interactive voice response system (IVRS) will be used to track subjects' assigned dose and study drug inventory. | | 7 |
| Section 9.4.6 Selection of Doses Used in the Study | The doses for this study will be based upon the results of findings in PAL-001 and PAL-002. | | 10 |
| Section 9.4.8 Prior and Concomitant Medications | Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and antihistamines and/or oral steroids (refer to Section 9.1.1). Subjects who have had a prior hypersensitivity reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and antihistamines and/or oral steroids (refer to Section 9.1.1). If the local or systemic reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study. | | 1 |
| 9.7.4.2 rAvPAL-PEG-<br>specific antibodies<br>Antibody Testing | Anti-PEG antibodies will also be measured. | Re-named section | 10 |

 February 09, 2009




| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| Section 14.3<br>Pharmacokinetic<br>Analysis | Should data become available from PAL-001 and/or PAL-002 which indicate study drug accumulation should also be measured, the protocol will be amended to require additional blood draws for PK analysis. | | 11 |
| Section 14.7 Interim<br>Analyses | At least one interim analysis may be performed by the sponsor during the study. | Added new section | 6 |



#### 2 SYNOPSIS

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

## TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

PROTOCOL NUMBER: PAL-003

**STUDY SITES:** Approximately 8 centers in the United States

PHASE OF DEVELOPMENT: Phase 2

#### STUDY RATIONALE:

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding study (Study PAL-002). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

## **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU who participated in Study PAL-002.
- To evaluate steady-state PK of rAvPAL-PEG in subjects with PKU.

| BIOMARIN | PAL-003 |
|----------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### STUDY DESIGN AND PLAN:

This is a long-term extension of a Phase 2, open-label, dose-finding study (Study PAL-002) in approximately 35 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002.

Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

A Data Monitoring Committee will monitor the study.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 participants' rAvPAL-PEG dosing will continue in PAL-003 without interruption of weekly dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations below 480 µmol/L. Subjects will continue to receive injections in the clinic, administered by clinic staff, but may later be allowed to self-administer doses of study drug at home. Whether a subject may be allowed to self-administer study drug doses will be evaluated on an individual basis.

The dose may be modified at any time for safety.

Evaluations, observations, and procedures will be conducted at selected timepoints as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been controlled to within a target range (below 480  $\mu$ mol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses.

A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The drug becomes commercially available following the appropriate marketing approval.
- 4. The study is terminated.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

# **Dose Adjustment Methodology:**

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Depending upon the response to rAvPAL-PEG in PAL-002, a subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- The dose may be decreased as appropriate to achieve or maintain a favorable blood Phe concentration.
- When adjusting the dose, a dose may be used that is between the dose cohort levels that were defined in the previous study (PAL-002).
- The dose may be adjusted by increasing the frequency of injections per week, up to one dose per day, for a maximum total dose per week of 2 mg/kg.
- When a dose is adjusted (either by changing the dose level or by changing the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time.

Subjects must have blood Phe concentration tested 3 days after a dose adjustment. There must be a minimum of 2 weeks after each dose adjustment before any additional dose adjustments may be made, so that blood Phe concentrations can be assessed.

# Stopping Criteria:

If an individual subject exhibits drug-related toxicity of CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level.

In addition, if 2 or more subjects at a dose level exhibit drug-related toxicity of CTCAE grade 3 or greater, further dosing of subjects at that dose level and any higher dose levels will be halted until a safety assessment is completed.

## NUMBER OF SUBJECTS PLANNED:

Approximately 35 subjects.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

## DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- Must have completed participation in PAL-002.
- Willing and able to provide written, signed informed consent, or, in the case of participants
  under the age of 18, provide written assent (if required) and written informed consent by a
  parent or legal guardian, after the nature of the study has been explained, and prior to any
  research-related procedures.
- Willing and able to comply with all study procedures.
- Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- Maintained a stable diet.
- In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
- Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

- A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product.
- Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL-001 or PAL-002.
- Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- Creatinine > 1.5 times the upper limit of normal.

# INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

rAvPAL-PEG doses will be administered SC and the favorable dose (the dosage that provides control of blood Phe concentrations within the target range for a minimum of 2 weeks) will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses.

## **DURATION OF TREATMENT:**

Extension of multiple dosing will continue until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The drug becomes commercially available following the appropriate marketing approval.
- 4. The study is terminated.



| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

#### **CRITERIA FOR EVALUATION:**

## **Efficacy:**

Blood Phe concentrations will be measured.

## **Safety:**

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs or laboratory test results.

#### **Pharmacokinetic:**

Plasma concentrations of rAvPAL-PEG will be measured when steady-state levels of Phe are attained.

## STATISTICAL METHODS:

## Sample Size:

Subjects who participated in PAL-002 may be enrolled into this study. No formal sample size calculation was conducted.

## **Safety Analysis:**

All subjects who receive any amount of study drug in this study will be included in the safety analyses.

Safety will be evaluated on the incidence of AEs, including serious AEs (SAEs), and clinically significant changes in vital signs and laboratory test results.

## **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any posttreatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled timepoint will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled timepoint will also be summarized.

#### **Pharmacokinetic Analysis:**

Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis.

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the



| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

subject has achieved and maintained target blood Phe concentration (below 480  $\mu$ mol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks.




## 2.1 Schedule of Events

**Table 2.1.1: Schedule of Events** 

| | Screening | | Treat | ment Period <sup>b,c</sup> | | Final F/U or<br>ETV |
|---|---|---|---|---|---|---|
| | | Week 1 | Weekly | Monthly (eg,<br>Wk 4, 8, etc, | Qrtly (eg,<br>Wk 12, 24,<br>etc) | 4 weeks after final dose |
| Assessments and Events | | D 1 | | | | |
| Informed consent | X | | | | | |
| Medical history and demographics | X | | | | | |
| Physical examination <sup>d</sup> | X | X | | | X | X |
| Vital signs | X | X | X | X | X | X |
| 12-lead ECG | X | | | | | X |
| Clinical laboratory tests <sup>e</sup> | X | | | X | X | X |
| Sedimentation rate | | X | | | X | X |
| Urine pregnancy test | X | X | | X | X | X |
| Injection-site inspectionf | | X<br>(postdose) | X | X | X | X |
| Adverse events <sup>g</sup> | Χ← | | | | | → X |
| Concomitant medications | X | X | X | X | X | X |
| Diet query | X | X | X | X | X | X |
| Serum rAvPAL-PEG antibodies | | X | | X | X | X |
| Predose blood Phe and plasma tyrosine <sup>h</sup> | X | X | X | X | X | X |
| Blood Phe (fingerstick) <sup>i</sup> | | | 3 days<br>postdos<br>e | | | |
| Predose PK sample <sup>j</sup> | | | | | | |
| Administer IP <sup>k</sup> | | X | X | X | X | |

AE, adverse event; D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> It is preferable to perform PAL-003 Screening assessments the same day as PAL-002 Final Follow-up Visit so there is no interruption of study drug. If performed on the same day, PAL-002 Final Follow-up Visit data may be used. If not, PAL-003 Day 1 must occur  $\leq$  28 days after PAL-003 Screening.

<sup>&</sup>lt;sup>b</sup> Additional visits may occur if deemed necessary to monitor AEs or blood Phe, adjust dosing etc.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Complete physical examinations to include the evaluation of all major body systems, height (at Screening only), and weight.



<sup>&</sup>lt;sup>e</sup> Clinical laboratory tests to include hematology, chemistry, and urinalysis.

- f If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, e.g. right arm vs. left arm)
- <sup>g</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug to the final study visit.
- <sup>h</sup> Samples should be drawn in the morning, at least 2.5 hours after a meal. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.
- <sup>1</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.
- j. The PK blood samples will be collected after the subject has achieved and maintained target blood Phe concentration (below 480 μmol/L) for a minimum of 2 weeks. Once this target is achieved, predose PK samples will be collected on the same day each week for 3 consecutive weeks as specified in Section 9.7.3.
- <sup>k</sup> Dosing is up to 1.0 mg/kg per injection and up to one dose per day, for a total of up to 2.0 mg/kg/week.




# **3 TABLE OF CONTENTS**

| 1 | TIT | LE PA | \GE | 1 |
|---|---|---|---|---|
| 2 | SYN | OPSIS. | | 16 |
| | 2.1 | | ule of Events | |
| 3 | TAB | | CONTENTS | |
| 4 | | | BBREVIATIONS AND DEFINITIONS OF TERMS | |
| 5 | | | | |
| J | 5.1 | | tional Review Board or Ethics Committee | |
| | 5.2 | | l Conduct of Study | |
| | 5.3 | | ct Information and Informed Consent | |
| 6 | | | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | |
| 7 | | | CTION | |
| , | 7.1 | | inical Studies | |
| | 7.2 | | ous Clinical Studies | |
| | 7.3 | | Rationale | |
| | 7.4 | | nary of Overall Risks and Benefits | |
| | , | 7.4.1 | Toxicity Due to Exposure to PEG | |
| | | 7.4.2 | | |
| | | | 7.4.2.1 Management of Allergic Reactions | |
| | | 7.4.3 | | |
| 8 | STII | , , , , , | BJECTIVES | |
| 9 | | | ATIONAL PLAN | |
| , | 9.1 | | ll Study Design and Plan | |
| | 7.1 | | Management of Local and Systemic Reactions to rAvPAL-PEG | |
| | | | 9.1.1.1 Subjects Who Have Experienced Hypersensitivity | |
| | | | Reactions to rAvPAL-PEG or a PEG-containing Product | 44 |
| | | 9.1.2 | Dose Adjustment Methodology | 47 |
| | | 9.1.3 | Stopping Criteria | |
| | 9.2 | Discus | ssion of Study Design, Including Choice of Control Group | |




| 9.3 | Selecti | on of Study Population | 48 |
|-----|---------|------------------------------------------------------|----|
| | 9.3.1 | Inclusion Criteria | 48 |
| | 9.3.2 | Exclusion Criteria | 48 |
| | 9.3.3 | Removal of Subjects from Treatment or Assessment | 49 |
| | 9.3.4 | Subject Identification and Replacement of Subjects | 50 |
| 9.4 | Treatm | nents | 50 |
| | 9.4.1 | Treatments Administered | 50 |
| | 9.4.2 | Identity of Investigational Product (IP) | 51 |
| | | 9.4.2.1 Product Characteristics and Labeling | 51 |
| | 9.4.3 | Storage | 51 |
| | 9.4.4 | Directions for Administration | 51 |
| | 9.4.5 | Method of Assigning Subjects to Treatment Groups | 52 |
| | 9.4.6 | Selection of Doses Used in the Study | 52 |
| | | 9.4.6.1 Selection of Timing of Dose for Each Subject | 53 |
| | 9.4.7 | Blinding | 53 |
| | 9.4.8 | Prior and Concomitant Medications | 53 |
| | 9.4.9 | Treatment Compliance | 54 |
| 9.5 | Investi | gational Product Accountability | 54 |
| | 9.5.1 | Return and Disposition of Clinical Supplies | 54 |
| 9.6 | Dietar | y or Other Protocol Restrictions | 54 |
| 9.7 | Efficac | cy and Safety Variables | 55 |
| | 9.7.1 | Efficacy and Safety Measurements Assessed | 55 |
| | | 9.7.1.1 Demographic Data and Medical History | 55 |
| | | 9.7.1.2 Physical Examination Findings | 55 |
| | | 9.7.1.3 Vital Sign Measurements | 55 |
| | | 9.7.1.4 Electrocardiography | 56 |
| | 9.7.2 | Efficacy Variable | 56 |
| | | 9.7.2.1 Blood Phenylalanine Concentrations | 56 |
| | 9.7.3 | Pharmacokinetic Variables | 56 |
| | 9.7.4 | Safety Variables | 56 |

| <b>B</b> OMARIN |
|-----------------|
|-----------------|


| | 9.7.4.1 Pregnancy Testing | 56 |
|---|---|---|
| | 9.7.4.2 Antibody Testing | 57 |
| | 9.7.5 Clinical Laboratory Assessments | 57 |
| 10 | REPORTING ADVERSE EVENTS | 59 |
| | 10.1 Adverse Events | 59 |
| | 10.2 Serious Adverse Events | 61 |
| | 10.3 Pregnancy | 62 |
| | 10.4 BioMarin Pharmacovigilance Contact Information | 62 |
| 11 | APPROPRIATENESS OF MEASUREMENTS | 63 |
| | 11.1 Pharmacokinetics | 63 |
| 12 | STUDY PROCEDURES | 64 |
| | 12.1 Prestudy | 64 |
| | 12.2 Screening Visit | 64 |
| | 12.3 Treatment Period | 65 |
| | 12.3.1 Day 1 (Week 1) | 65 |
| | 12.3.2 Weekly Visits | 66 |
| | 12.3.3 Monthly Visits (Week 4, 8, 16, etc) | 66 |
| | 12.3.4 Quarterly Visits (Week 12, 24, 36, etc) | 67 |
| | 12.4 Final Follow-up Visit (Day 113 [± 3 days]) /Early Termination Visit | 68 |
| 13 | DATA QUALITY ASSURANCE | 69 |
| 14 | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 70 |
| | 14.1 Statistical and Analytical Plans | 70 |
| | 14.2 Safety Analysis | 70 |
| | 14.3 Pharmacokinetic Analysis | 70 |
| | 14.4 Efficacy Analysis | 70 |
| | 14.5 Determination of Sample Size | 71 |
| | 14.6 Handling of Missing Data | 71 |
| | 14.7 Interim Analyses | 71 |
| | 14.8 Changes in the Conduct of the Study or Planned Analyses | 71 |
| 15 | DATA MONITORING COMMITTEE (DMC) | 72 |

| BIOMARIN | PAL-003 | |
|---|---|---|
| 16 COMPENSATION, INS | SURANCE, AND INDEMNITY | 73 |
| 17 CASE REPORT FORM | IS AND SOURCE DOCUMENTS | 74 |
| 18 STUDY MONITORING | G AND AUDITING | 76 |
| 19 RETENTION OF RECO | ORDS | 77 |
| 20 USE OF INFORMATION | ON AND PUBLICATION | 78 |
| 21 REFERENCES | | 79 |
| 22 INVESTIGATOR RES | PONSIBILITIES | 81 |
| 22.1 Conduct of Study | and Protection of Human Subjects | 81 |
| LIST OF TABLES | | |
| Table 2.1.1: Schedule of Ex | vents | 23 |
| Table 9.4.4.1 Number of In | jections Required For an Individual W | Teighing 80 kg52 |
| Table 9.7.1.1: Summary of | Laboratory Assessments | 55 |
| Table 9.7.5.1: Clinical Laboratory | pratory Tests | 58 |
| LIST OF FIGURES | | |

Figure 9.1.1.1.2.1: Management of Local and Systemic Reactions to rAvPAL-PEG......46




## 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

 $AUC_{0-7\;days}$  area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen

°C degree Celsius

C<sub>trough</sub> predose concentration of rAvPAL-PEG

CD Compact disk

CFR Code of Federal Regulations

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form

CTCAE Common Terminal Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure
DCF Data Clarification Form

DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

f/u follow-up

g gram

GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure

| B <u>!</u> OMARIN | PAL-003 |
|-------------------|---------|

ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IgG immunoglobulin G IgM immunoglobulin M

IND Investigational New Drug
IP investigational product
IRB Institutional Review Board

IV intravenous

IVRS interactive voice response system

kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

NAb neutralizing antibodies

NCI National Cancer Institute

OTC over the counter

PAH phenylalanine hydroxylase PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator
PK pharmacokinetics
PKU phenylketonuria

rAvPAL-PEG phenylalanine ammonia lyase

RBC red blood cell

SAE serious adverse event
SAP Statistical Analysis Plan
SBP systolic blood pressure

SC subcutaneous

SD standard deviation SDV source data verified

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

SGOT serum glutamic oxalo-acetic transaminase SGPT serum glutamic pyruvate transaminase

US United States
WBC white blood cell



# Definition of Terms:

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.



## 5 ETHICS

# 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

# 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will



provide written, informed consent before any study-related tests or evaluations are performed.

# 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR §50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



## 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Regulatory Affairs Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.




## 7 INTRODUCTION

A comprehensive review of phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

# 7.1 Nonclinical Studies

The murine model of phenylketonuria (PKU) BTBRPah<sup>enu2</sup> (ENU<sup>2</sup>), a mouse line that is deficient in phenylalanine hydroxylase (PAH) activity (Shedlovsky, 1993, Genetics), was used for in vivo screening and pharmacodynamic studies. This mouse model exhibits characteristics similar to those seen in PKU patients, including hyperphenylalaninemia (baseline plasma phenylalanine [Phe] concentrations of 1000 to 2000 µM) and hypopigmentation. Weekly subcutaneous (SC) administration of 80 mg/kg of rAvPAL-PEG (approximately 4 IU/mouse) for greater than 3 months lowered blood Phe concentration from approximately 2000 μM to less than 200 μM. A similar profile of Phe reduction was also seen in ENU<sup>2</sup> mice administered wild-type AvPAL-PEG (4 IU/mouse) over 8 weeks. In all these studies, regardless of the molecule, an attenuated Phe-lowering response was usually seen between Weeks 2 and 7. However, plasma Phe concentrations became stabilized at concentrations below 200 µM from Week 7 onward. In addition to the reduction of plasma Phe, a dose-related darkening in coat color occurred, indicating the biosynthesis of melanin, which was previously inhibited when plasma Phe could not be metabolized and plasma Phe concentrations were high. When administration of AvPAL-PEG was stopped for 2 to 7 weeks and then reinitiated with weekly administrations, no attenuated response was observed and Phe concentrations remained low and stable until the next administration.

The safety of rAvPAL-PEG was evaluated in safety pharmacology studies (respiratory, central nervous system [CNS] and cardiovascular [CV]) and toxicity with toxicokinetic studies (single and 28-day repeated dose) in rats and cynomolgus monkeys. Overall, in all toxicity studies no immune-related toxicities were seen either systemically or at the injection site. No specific polyethylene glycol (PEG)-related histological findings were observed during the 28-day repeated dose studies.

Findings in cynomolgus monkeys dosed with a single administration of 60 mg/kg rAvPAL-PEG included **reduced food consumption**, **dehydration**, **body weight loss**, **hypoactivity**, **hypothermia**, decreased plasma Phe concentration, decreased protein synthesis, and gastrointestinal (GI) lesions. Plasma Phe concentrations were also reduced to below the level of detection in the 4 and 12 mg/kg dose groups, but without similar




toxicological consequence, implying that the physiological regulation of Phe levels may be an important factor for influencing morbidity.

The main finding in the 28-day study was the possible drug-related observation of minimal to slight degeneration of blood vessels of predominantly medium-sized muscular arteries with a non-dose-dependent involvement of different organs observed in 1 male in the 0.1 mg/kg and 1 male and 1 female in the 1.0 mg/kg rAvPAL-PEG dose groups. No degeneration of the arteries was observed in animals administered 0 and 0.01 mg/kg rAvPAL-PEG.

The half-life of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg, was 47, 33, and 44 hours, respectively, and exhibited modest area under the plasma concentration-time curve (AUC)-dose linearity. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the half-life was 65 hours at 4 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum plasma concentration, along with a long half-life, (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) AUC and the maximum plasma concentration (C<sub>max</sub>) are roughly linearly proportional.

## 7.2 Previous Clinical Studies

This study is an extension of the second human clinical study with rAvPAL-PEG (Study PAL-002). Study PAL-001, the first-in-human clinical study of rAvPAL-PEG, was designed as a Phase 1, open-label, single-dose, dose-escalation study in approximately 35 subjects, 16 to 50 years old, with PKU. The doses for this study are planned to be in the same range as those tested in PAL-001 and PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in those studies.

# 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH (Scriver CR, 2001, McGraw-Hill). Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver CR, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and




behavioral abnormalities (Scriver CR, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Leey, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan® is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding study (PAL-002). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

# 7.4 Summary of Overall Risks and Benefits

It is not expected that data from PAL-001 and PAL-002 will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.




# 7.4.1 Toxicity Due to Exposure to PEG

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given up to 60 mg/kg of SC rAvPAL-PEG.

In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

# 7.4.2 Toxicity Due to an Immunologic Reaction

The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. In animal models, the immune response against the foreign protein PAL in rAvPAL-PEG has been mitigated by PEGylation. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylation does not eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing the immunogenicity of the molecule, it is reasonable to expect that some individuals may exhibit immune responses upon exposure to the drug. These immune responses may be clinically irrelevant, cause symptoms of various degrees, or lead to neutralization of biological activity. Subjects participating in clinical trials will be monitored closely with specific antibody titers, sedimentation rates, and complete blood counts (CBCs).

PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.) (Harris, 2003, Nat.Rev.Drug Discov.), however, antibodies against PEG may form when PEG is bound to compounds. (Harris, 2003, Nat.Rev.Drug.Discov.) (Richter, 1983, Int.Arch.Allergy Appl.Immunol.) In some instances, development of such antibodies did not result in any significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.).

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

Two subjects enrolled in PAL-001 who had received one dose of rAvPAL-PEG experienced hypersensitivity reactions to intramuscular (IM) Depo-Provera, a contraceptive containing PEG 3350. Both subjects had previously received multiple IM Depo-Provera injections without complications.



Because Depo-Provera contains PEG 3350 as an excipient, it is possible that the administration of rAvPAL-PEG caused anti-PEG antibody formation that led to a cross-reaction with Depo-Provera in these subjects. Therefore, it is possible that prior exposure to rAvPAL-PEG might sensitize subjects to other PEG-containing injectable drugs. Alternatively, the presence of Depo-Provera could have led to antibody formation and cross-reaction with rAvPAL-PEG, leading to rAvPAL-PEG injection-site reactions. Since it is currently unknown whether Depo-Provera has a sensitizing effect to PEG and the exact basis for these reported events is not known, the use of PEG-containing injectable drugs prior to and during the study is prohibited as a precautionary measure (refer to the addendum and Sections 9.3.2 and 9.4.8).

Allergic reactions to the SC injection of rAvPAL-PEG may be mild, moderate or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or




anaphylaxis. Clinical assessments should be conducted for a minimum of 2 hours post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of allergic reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection.

In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for antibody testing. This additional testing may occur up to 6 months following the final study visit.

# 7.4.2.1 Management of Allergic Reactions

The following measures are recommended for the treatment of allergic symptoms:

- Clearing the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. Acetaminophen or ibuprofen (5-10 mg/kg) may also be administered. An allergy and/or immunology consultation should be sought if necessary.

## 7.4.3 Effects of Low Blood Phe

Insufficient Phe intake or excessive rAvPAL-PEG exposure may cause blood Phe concentrations to be too low (eg, < 30 °m ol/L). Prolonged low blood Phe concentrations can result in a catabolic state associated with poor growth and altered body functions, including mental and physical alterations, loss of appetite, anemia, rashes, and diarrhea. To ensure safety during this study, subjects will be monitored closely with frequent blood Phe concentration determinations.



# 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU who participated in Study PAL-002.
- To evaluate steady-state PK of rAvPAL-PEG in subjects with PKU.



## 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of a Phase 2, open-label, dose-finding study (PAL-002) in approximately 35 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002.

Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

A Data Monitoring Committee will monitor the study.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 participants' rAvPAL-PEG dosing will continue in PAL-003 without interruption of weekly dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations below 480 µmol/L based upon recommendations by the German Working Group for Metabolic Diseases (Burgard, 1999, Eur J Pediatr). Subjects will continue to receive injections in the clinic, administered by clinic staff, but may later be allowed to self-administer doses of study drug at home. Whether a subject may be allowed to self-administer study drug doses will be evaluated on an individual basis. All of the following criteria must be met before a subject may self-administer doses of the study drug:

- The subject is willing and able to administer the study drug as directed.
- The sponsor agrees that self-administration is appropriate.
- The subject has achieved a favorable dose (ie, the dosage that provides control of blood Phe concentrations within the target range for a minimum of 2 weeks).
- The subject has received appropriate training, including administering doses under supervision, until the subject and clinic staff both agree such training is no longer necessary.

The dose may be modified at any time for safety.

Evaluations, observations, and procedures will be conducted at selected timepoints as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been



controlled to within a target range (below 480 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses.

A subject will continue in PAL-003 until one of the following occurs:

- 12. The subject withdraws consent and discontinues from the study.
- 13. The subject is discontinued from the study at the discretion of the Investigator.
- 14. The drug becomes commercially available following the appropriate marketing approval.
- 15. The study is terminated.

# 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEG

# 9.1.1.1 Subjects Who Have Experienced Hypersensitivity Reactions to rAvPAL-PEG or a PEG-containing Product

Subjects who had a previous reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from PAL-001 or PAL-002 are excluded from this study. However, subjects may develop such reactions after enrollment in PAL-003. Management of such reactions are described below. Refer to Figure 9.1.1.1.2.1 for a flowchart for managing these subjects.

# 9.1.1.1.1 Subjects with Local Reactions

After enrollment in PAL-003, subjects who have a local reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophpen and antihistamines and/or oral steroids, 1 hour prior to study drug dosing. Recommended premedications are acetaminophen and antihistamine (Claritin is preferred). The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg Claritin or 25 to 50 mg oral Benadryl; an example for steroids would be 70 mg oral prednisone). Because Benadryl can cause drowsiness, it should be administered only if the subject is accompanied by a designated driver.

# 9.1.1.1.2 Subjects with Systemic Reactions

After enrollment in PAL-003, subjects who have a systemic reaction that includes noncutaneous systemic symptoms, such as respiratory problems, hypotension, or angioedema, to rAvPAL-PEG or a PEG-containing product will be evaluated with a skin prick test. If the test is positive, the subject will be excluded from the study.



Subjects with prior systemic reactions that included only skin manifestations to rAvPAL-PEG or a PEG-containing product after PAL-003 enrollment will be premedicated with acetaminophen and antihistamines and/or oral steroids (one hour prior to study drug dosing) and will continue to receive rAvPAL-PEG.

Reactions to skin prick testing or rAvPAL-PEG administered SC are defined as follows:

<u>Local reaction</u>: 1 affected location, ie, hives, wheals, or swelling or an area of erythema or redness at or near the site of injection.

<u>Systemic reaction</u>: more than 1 affected location, ie, cutaneous reaction in more than 1 area, and/or any other generalized symptoms, such as hypotension, angioedema or anaphylaxis or the involvement of other organ systems (eg, respiratory, cardiovascular, gastrointestinal).


Figure 9.1.1.1.2.1: Management of Local and Systemic Reactions to rAvPAL-PEG





#### 9.1.2 Dose Adjustment Methodology

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Depending upon the response to rAvPAL-PEG in PAL-002, a subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- The dose may be decreased as appropriate to achieve or maintain a favorable blood Phe concentration.
- When adjusting the dose, a dose may be used that is between the dose cohort levels that were defined in the previous study (PAL-002).
- The dose may be adjusted by increasing the frequency of injections per week, up to one dose per day, for a maximum total dose of 2 mg/kg/week.
- When a dose is adjusted (either by changing the dose level or by changing the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time.

Subjects must have blood Phe concentration tested 3 days after a dose adjustment. There must be a minimum of 2 weeks after each dose adjustment before any additional dose adjustments may be made so that blood Phe concentrations can be assessed.

## 9.1.3 Stopping Criteria

If an individual subject exhibits drug-related toxicity of CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principle Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level.

In addition, if 2 or more subjects at a dose level exhibit drug-related toxicity of CTCAE grade 3 or greater, further dosing of subjects at that dose level and any higher dose levels will be halted until a safety assessment is completed.

## 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.



## 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- Must have completed participation in PAL-002.
- Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- Willing and able to comply with all study procedures.
- Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- Maintained a stable diet.
- In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

#### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product.
- Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.




- Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- Creatinine > 1.5 times the upper limit of normal.

# 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study at any time without prejudice. The Investigator must withdraw from the study any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject experiences a serious or intolerable AE.
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).



If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

# 9.3.4 Subject Identification and Replacement of Subjects

Each subject was assigned a unique subject identifier in either PAL-001 or PAL-002. Subjects will retain the same subject number used in PAL-002.

This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

After enrollment of 35 subjects, if any single cohort (identified during PAL-002) has less than 3 subjects due to early terminations, those subjects will be replaced. Replacement subjects will enter the study at the same dose cohort level as the subject they are replacing.

#### 9.4 Treatments

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site with a supply of IP sufficient for the completion of the study.




#### 9.4.2 Identity of Investigational Product (IP)

# 9.4.2.1 Product Characteristics and Labeling

The rAvPAL-PEG drug product for SC injection is formulated and supplied as a sterile aqueous (colorless to pale yellow) solution in clear, single-use, type-1 borosilicate glass vials. Each 3 mL vial contains  $1.5\pm0.2$  mL to deliver 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with  $1.5\pm0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Dilution instructions are provided in a separate instruction manual.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

Drug product packaging will be identified with the lot number and expiration date, and will be provided in a box labeled with the study number.

## 9.4.3 Storage

At the study site, all IP must be stored at  $5\pm3^{\circ}$ C ( $41\pm5^{\circ}$ F) under the conditions specified in the IB in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 2 mg/kg.

Dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

The injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper



arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). The number of injections required for an individual weighing 80 kg (about 176 pounds) is provided in Table 9.4.4.1 as an example, Note this table is for example purposes only. Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual.

Table 9.4.4.1 Number of Injections Required For an Individual Weighing 80 kg

| Dose Group<br>(mg/kg) | Weight (kg) | Volume of Study Drug (mL) <sup>a</sup> | No. of<br>Injections <sup>b</sup> |
|---|---|---|---|
| 0.001 | 80 | 0.8 | 1 |
| 0.003 | 80 | 0.6 | 1 |
| 0.01 | 80 | 0.8 | 1 |
| 0.03 | 80 | 0.2 | 1 |
| 0.1 | 80 | 0.8 | 1 |
| 0.3 | 80 | 2.4 | 2 |
| 1.0 | 80 | 8.0 | 4 |

<sup>&</sup>lt;sup>a</sup>Study drug is supplied at a concentration of 10 mg/mL and is then diluted by differential amounts as specified in the PAL-003 Pharmacy Manual. Volume to be injected is calculated based on a starting volume attained following dilution.

# 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in PAL-002.

An interactive voice response system (IVRS) will be used to track subjects' assigned dose and study drug inventory.

#### 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU.

<sup>&</sup>lt;sup>b</sup>Number of injections per dose is dependent upon site policy for SC injections. The number of injections may vary at the discretion of the Investigator.




A favorable dose that produces a reduction in blood Phe concentration to below 480  $\mu$ mol/L will be determined for each subject. Findings in cynomolgus monkeys dosed with a single administration of 60 mg/kg rAvPAL-PEG included severe morbidity, decreased plasma Phe concentration, decreased protein synthesis, and GI lesions. Plasma Phe concentrations were reduced to below the level of detection in the lower dose groups, without other findings. The doses for this study will be based upon the **findings in** PAL-001 and PAL-002.

## 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered in the morning by clinic staff or by the subject, if appropriate.

## 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the medical monitor must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in PAL-002) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and antihistamines and/or oral steroids (refer to Section 9.1.1).

Subjects who have had a prior hypersensitivity reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and antihistamines and/or oral steroids (refer to Section 9.1.1). If the local or systemic reaction worsens with a repeat injection (as determined by the Investigator in consultation with the




# Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study.

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

# 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

# 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

# 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

# 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study except as necessary for safety.



## 9.7 Efficacy and Safety Variables

## 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis (Section 2.1) describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

**Table 9.7.1.1: Summary of Laboratory Assessments** 

| <b>Laboratory Assessment</b> | Party Responsible for<br>Performing Test | Section in Protocol for Details |
|---|---|---|
| Clinical laboratory tests | Central laboratory | 9.7.5 |
| Antibody testing | BioMarin | 9.7.4.2 |
| PK variables | Central laboratory | 9.7.3 |
| Blood Phe concentrations | Central laboratory | 9.7.2.1 |

Phe, phenylalanine; PK, pharmacokinetic.

## 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

#### 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of weight; general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Height will be measured at Screening only. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

#### 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury



(mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C).

## 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the final follow-up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

## 9.7.2 Efficacy Variable

# 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn in the morning, at least 2.5 hours after a meal, on the days and timepoints indicated in the Schedule of Events (Table 2.1.1).

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 480 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks.

BioMarin will perform the analysis.

## 9.7.4 Safety Variables

## 9.7.4.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the timepoints specified in the Schedules of Events (Table 2.1.1). Female subjects with a positive pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test results.



Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

## 9.7.4.2 Antibody Testing

Immunoglobulin G (IgG) and M (IgM) antibodies and neutralizing antibodies (NAb) to rAvPAL-PEG will be measured using validated immunogenicity assays at the timepoints indicated in the Schedule of Events (Table 2.1.1). **Anti-PEG antibodies will also be measured.** 

BioMarin will perform the analysis.

# 9.7.5 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.

Specific days for obtaining samples are provided in Table 2.1.1 and in Section 12. The scheduled clinical laboratory tests are listed in Table 9.7.5.1. A central laboratory will be used for analysis.




**Table 9.7.5.1: Clinical Laboratory Tests** 

| <b>Blood Chemistry</b> | Hematology | <b>Urine Tests</b> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if applicable |
| Alkaline<br>Phosphatase | Hematocrit | Color | |
| ALT (SGPT) | WBC count | pН | Pharmacokinetics |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Serum rAvPAL-PEG-<br>specific antibodies<br>(IgG, IgM, and NAb) |
| BUN | Differential cell count | Protein | |
| Creatinine | Sedimentation rate | Glucose | |
| GGT | | Bilirubin | Phenylalanine |
| Total protein | | Nitrite | |
| Calcium | | Urobilinogen | |
| Sodium | | Hemoglobin | |
| Potassium | | | |
| Glucose | | | |
| Uric acid | | | |
| CO <sub>2</sub> | | | |
| Chloride | | | |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; CO<sub>2</sub>, carbon dioxide; GGT, gamma-glutamyltransferase; IgG, immunoglobulin G; IgM, immunoglobulin M; NAb, neutralizing antibodies; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.



#### 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

According to the ICH definition, an AE (or adverse experience) is "any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the IP."

An adverse drug reaction (ADR) is described by the ICH as "all noxious and unintended responses to a medicinal product related to any dose." This means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility, ie, the relationship cannot be ruled out.

An AE may include intercurrent illnesses or injuries that represent an exacerbation (increase in frequency, severity, or specificity) of pre-existing conditions (eg, worsening of asthma). Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The reporting period for non-serious AEs is the period from the first administration of study drug through the final F/U Visit or at the ETV. If a non-serious AE remains unresolved at the conclusion of the study, the PI and medical monitor will make a joint clinical assessment as to whether continued follow-up of the AE is warranted, and the results of this assessment must be documented. Resolution is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

The Investigator will assess AEs for severity, for relationship to IP, and as to whether the event meets one or more of the definitions of an SAE (refer to Section 10.2).

The Investigator will determine the severity of each AE and will record it on the source documents and AE CRF, using the categories defined below.

| Grade | Description |
|----------|-----------------------------------------|
| Mild | No limitation of usual activities |
| Moderate | Some limitation of usual activities |
| Severe | Inability to carry out usual activities |



The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as "serious," which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the relationship of an AE to the IP and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably<br>Related | The administration of IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE is more likely explained by exposure to the IP than by other |
| | factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).



#### **10.2** Serious Adverse Events

A SAE is defined as any AE that:

- Results in death.
- Is life threatening, that is, places the subject at immediate risk of death from the event as it occurred. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires in-patient hospitalization or prolongation of an existing in-patient hospitalization. Admission of a subject to the hospital as an in-patient as a result of an AE, even if the subject is released on the same day, qualifies as hospitalization.
- Results in persistent or significant disability or incapacity. An event qualifies as
  resulting in a persistent or significant disability or incapacity if it involves a
  substantial disruption of the subject's ability to carry out usual life functions.
  This definition is not intended to include experiences of relatively minor or temporary
  medical significance.
- Is a congenital anomaly or birth defect, that is, an AE that occurs in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Is an important medical event that does not meet any of the above criteria, but may jeopardize the subject or require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such events are intensive treatment in the emergency room, allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

More than one of the above criteria may apply to any specific event.

The reporting period for SAEs begins earlier than non-serious AEs and is the period from the time of signing of the ICF through 4 weeks after the last dose or at the ETV. SAEs reported to the Investigator outside of this reporting period will be reported to BioMarin if, in good medical judgment, the event has any bearing on the study data. SAEs must be followed by the Investigator until resolution, even if this extends beyond the study-reporting period. Resolution of an SAE is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

Any SAE, whether or not considered related to study drug, will be reported immediately (within 24 hours) to BioMarin Pharmacovigilance by fax using the study-specific SAE Report Form. In addition to the outcome of the SAE, any medication or other therapeutic measures used to treat the event will be recorded on the appropriate CRF page(s). Investigators should not wait to collect additional information that fully documents the event before notifying BioMarin Pharmacovigilance of an SAE. BioMarin may be required to




report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit additional information requested by BioMarin as soon as it becomes available.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

# 10.3 Pregnancy

Pregnancy in a subject or partner should be reported immediately (within 24 hours) to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up Form in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

## 10.4 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the medical monitor any AEs for which the issue of seriousness is unclear or questioned. Contact information for the medical monitor is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:

Fax: E-mail:


February 09, 2009



## 11 APPROPRIATENESS OF MEASUREMENTS

## 11.1 Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.



#### 12 STUDY PROCEDURES

## 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

# 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history and demographics
- Physical examination and height
- Vital signs
- 12-lead ECG
- Clinical laboratory tests (including hematology, chemistry, and urinalysis)
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration

For subjects who participated in PAL-002, these assessments may be the same used for the Final Follow-up Visit of PAL-002, if they occur within 28 days from Day 1.



#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done on the third day following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

## 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (postdose)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)



#### 12.3.2 Weekly Visits

The following study activities will be performed at the weekly visits beginning with Week 2:

- Vital signs
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasm tyrosine concentration
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

## 12.3.3 Monthly Visits (Week 4, 8, 16, etc)

The following study activities will be performed at the monthly visits beginning with Week 4:

- Vital signs
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)



## 12.3.4 Quarterly Visits (Week 12, 24, 36, etc)

Quarterly visits consist of all monthly activities and include additional activities. The following study activities will be performed at the quarterly visits beginning with Week 12:

- Physical examination
- Vital signs
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)




## 12.4 Final Follow-up Visit (Day 113 [± 3 days]) /Early Termination Visit

The final follow-up (F/U) Visit or Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the F/U Visit or ETV:

- Physical examination and weight
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies



## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.




#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

## 14.2 Safety Analysis

All subjects who receive any amount of study drug will be included in the safety analyses.

Safety will be evaluated on the incidence of AEs and clinically significant changes in vital signs and laboratory test results.

The verbatim terms reported on CRFs to identify AEs will be coded using MedDRA. Treatment-emergent AEs will be summarized for each treatment group by system organ class, preferred term, relationship to study drug, and severity. Changes from baseline in vital signs and laboratory test results will be summarized with descriptive statistics by dose group.

## 14.3 Pharmacokinetic Analysis

Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis.

Steady-state PK of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 480  $\mu$ mol/L) for a minimum of 2 weeks and no further dose modification is planned.

Should data become available from PAL-001 and/or PAL-002 which indicate study drug accumulation should also be measured, the protocol will be amended to require additional blood draws for PK analysis.

## 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any posttreatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled timepoint will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration



from baseline to each scheduled timepoint and presence/absence of antibodies will also be summarized.

## 14.5 Determination of Sample Size

Subjects who participated in PAL-002 may be enrolled into this study. No formal sample size calculation was conducted.

# 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.

## 14.7 Interim Analyses

At least one interim analysis may be performed by the sponsor during the study.

## 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.



## 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act in an advisory capacity to BioMarin to monitor subject safety and the efficacy of rAvPAL-PEG in subjects who participate in the study. Meetings of the DMC can be convened at any time at the discretion of the DMC Chair or the Study Medical Officer. The Chair will be notified by the Study Medical Officer of all SAEs and will receive summaries of other safety data as available. The DMC will review the study data as soon as it is available during the study, on a schedule defined in the DMC Charter, and offer advice on whether or not to proceed, modify or terminate study enrollment on the basis of toxicity. Details regarding the DMC membership and safety data to be reviewed by members will be provided in a charter.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.3.



## 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment. If the subject has followed the Investigator's instructions, BioMarin will pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures, if these costs are not covered by health insurance or another third party that usually pays these costs. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.




#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent. If an Investigator or institution refuses to allow access to subject records because of confidentiality, arrangements must be made to allow an "interview" style of data verification.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.



#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (eg, subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.



## 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.




#### 21 REFERENCES

Armstrong, Hempel, Koling, Chan, Fisher, Meiselman, Garratty. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007.

Burgard, Bremer, Bührdel, Clemens, Mönch, Przyrembel, Trefz, Ullrich. Rationale for the German recommendations for phenylalanine level control in phenylketonuria 1997. Eur J Pediatr 158, 46-54. 1999.

Butterworth. Effects of hyperammonaemia on brain function. J Inherit Metab Dis 21 Suppl 1, 6-20. 1998.

Chen, Scott. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001.

Davis, Abuchowski, Park, Davis. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981.

Fisch. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000.

Gamez, Wang, Sarkissian, Wendt, Fitzpatrick, Lemontt, Scriver, Stevens. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007.

Ganson, Kelly, Scarlett, Sundy, Hershfield. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006.

Guttler, Azen, Guldberg, Romstad, Hanley, Levy, Matalon, Rouse, Trefz, de la, Koch. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003.

Harris, Chess. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003.

Huttenlocher. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000.

Kaufman. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989.




Koch, Hanley, Levy, Matalon, Matalon, Rouse, Trefz, Guttler, Azen, Platt, Waisbren, Widaman, Ning, Friedman, de la. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003.

Lee, Lilburn, Baudin. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003.

Levy. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003.

Matalon, Surendran, Matalon, Tyring, Quast, Jinga, Ezell, Szucs. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003.

Richter, Akerblom. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983.

Richter, Akerblom. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984.

Rouse, Azen. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004.

Scott, Murad, Koumpouras, Talbot, Eaton. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997.

Scriver CR, Kaufman S. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-709.

Shedlovsky, McDonald, Symula, Dove. Mouse models of human phenylketonuria. Genetics 134[4], 1205-1210. 1993.

Walter, White, Hall, MacDonald, Rylance, Boneh, Francis, Shortland, Schmidt, Vail. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002.

Webster, Didier, Harris, Siegel, Stadler, Tilbury, Smith. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007.



#### 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.


## 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

| Investigator Signature | Date |
|------------------------|------|
| Printed name: | |

# Accepted for the Sponsor:

On behalf of BioMarin, I confirm that BioMarin, as a sponsor will comply with all obligations as detailed in all applicable regulations and guidelines. I will ensure that the PI is informed of all relevant information that becomes available during the conduct of this study.

| | 2 | 118/09 |
|---------------|---|--------|
| | | Date |
| Printed name: | | |



#### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Study Title: Long-term Extension of a Phase 2, Open-Label Dose-Finding

> Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with

**PKU** 

**Protocol Number:** PAL-003

**Investigational Product:** rAvPAL-PEG IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria

BioMarin Pharmaceutical Inc. Sponsor:

> 105 Digital Drive Novato, CA 94949

**Development Phase:** Phase 2

Sponsor's Responsible

, MD Medical Officer:

Clinical Sciences

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

**Duration:** 24 months or until study is terminated

0.001 to 1.0 mg/kg per individual injection, with a maximum Dose:

weekly dose of 2.0 mg/kg

October 08, 2008 **Date of Original Protocol:** 

Date of Amendment 1: February 09, 2009 Date of Amendment 2: October 30, 2009

## **Property of BioMarin** CONFIDENTIAL

May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.



#### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

**Amendment: 2** 

Date: October 30, 2009

### RATIONALE AND SUMMARY OF CHANGES

- 1. The primary objective of the study has been revised for clarity; multiple doses of SC injections of rAvPAL-PEG will be assessed for efficacy on blood Phe levels of subjects with phenylketonuria (PKU).
- 2. Information regarding study drug dose adjustment (ie, allowable dose increases to achieve target Phe concentrations [ie, 120-600 μmol/L] and dose de-escalation for safety [ie, Phe concentration <120 μmol/L]) have been revised for clarity. Information regarding dose decreases relative to changes to subject diet has also been clarified.
- 3. Additional pharmacokinetic (PK) sampling has been added to allow for additional assessment of study drug exposure and accumulation based on PK information from the Phase 1 study, PAL-001 (A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single, Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria).
- 4. The information regarding the 2 subjects who reported serious adverse events in Study PAL-001 (A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single, Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria) has been updated. In addition, information regarding the future risk of using other PEG-containing or PEGylated injectable drugs has been added.
- 5. The Nonclinical Studies section has been updated to include information regarding chronic repeat-dose toxicity and toxicokinetic studies in monkeys and rats.
- 6. The stopping criteria have been revised for clarity.
  - The criterion for toxicity has been clarified; subjects who have a drug-related Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 event that is treatment emergent will stop study drug until resolution of the event.

|----------|---------|--------|
|----------|---------|--------|

- The criterion for stopping dosing within a dose level has been clarified; if 2 or more subjects within a dose level have a drug-related CTCAE grade ≥3 event that is treatment emergent, further dosing within that dose level will be stopped and no subjects in higher dose levels will be treated until a safety assessment is completed. The Food and Drug Administration (FDA) will also be notified.
- 7. Information regarding the management of local and systemic reactions to rAvPAL-PEG has been revised for clarity and to incorporate safety measures based on information from the Phase 1 study, PAL-001, and recommendations from an allergy advisory board.
  - The definition of local skin reactions (at or near the injection site) has been revised for further clarity.
  - Definitions of large local skin reactions that are contiguous and are not contiguous to the study drug injection site have been added.
  - The definition of systemic reactions has been revised to include skin (eg, generalized skin reaction) and non-skin symptoms; the definition has also been broadened for further clarity. In addition, the skin prick test for subjects with systemic reactions has been removed.
  - Information regarding subjects who have a systemic reaction that includes skin symptoms (eg, generalized skin reaction) has been revised. Subjects who have a generalized skin reaction will complete an Unscheduled Hypersensitivity Reaction Visit and will then be terminated from the study.
- 8. An Unscheduled Hypersensitivity Reaction Visit has been added for subjects who have a systemic reaction that includes skin symptoms (eg, generalized skin reaction) after administration of rAvPAL-PEG based on additional safety information from the Phase 1 study, PAL-001, and per the recommendation of an allergy advisory board.
  - The Unscheduled Hypersensitivity Reaction Visit includes clinical laboratory tests (urinalysis, hematology, chemistry) and tests for C-reactive protein (CRP), total hemolytic complement (CH50), complements C<sub>1</sub> and C<sub>4</sub>, sedimentation rate, serum tryptase level, and serum anti-rAvPAL-PEG antibodies to be performed within 48 hours of the reaction. A PK sample will also be obtained.
  - Subjects who have a large local skin reaction that is not contiguous to the injection site and subjects who have a systemic reaction that does not include skin symptoms (generalized skin reaction) may also have the Unscheduled Hypersensitivity Reaction Visit assessments performed per Investigator discretion and in consultation with the Sponsor's Medical Officer.

|----------|---------|--------|
|----------|---------|--------|

- All subjects who complete an Unscheduled Hypersensitivity Reaction Visit will be terminated from the study and will complete the Early Termination Visit assessments.
- 9. Information regarding treatment of subjects with local skin reactions has been revised to incorporate recommendations made by an allergy advisory board.
  - For subjects who have had a prior local skin reaction to rAvPAL-PEG or PEG-containing product, pretreatment with oral steroids has been removed because long-term steroid use is not indicated for the study patient population. The preferred antihistamine has been changed from Claritin (loratadine) to Zyrtec (cetirizine).
  - Information regarding treatment of subjects who have a local skin reaction has been added. Subjects may be treated with non-sedating oral and/or topical antihistamines and/or topical steroids.
- 10. Safety, PK, and blood Phe concentration assessments have been added for subjects who have their dose of rAvPAL-PEG increased in frequency to more than 1x/week. Subjects who have study drug frequency increased to 2x/week or daily should perform the Interim Dosing Visit assessments.
- 11. Dosing information has been revised to incorporate the additional dose levels in PAL-002. In addition, information regarding self-administration of study drug by subjects has been removed; study drug will be administered by the study clinic staff or other qualified and trained study personnel only.
- 12. Information regarding missed doses has been added. Subjects who miss more than 2 scheduled doses will need to have their dose level and dose frequency re-evaluated.
- 13. Information regarding the number of enrolled subjects has been revised to incorporate changes to Study PAL-002. In addition, information regarding replacement of subjects who do not complete the study has been removed. Only subjects who complete Study PAL-002 are eligible for participation in this study.
- 14. Information regarding assessment for immunogenicity has been clarified; the specific antibody assessments have been clarified per FDA request.
- 15. A 3-day diet diary has been added to the weekly visits.
- 16. The severity grades for adverse event (AE) reporting have been revised; CTCAE grades 1-5 will now be used.
- 17. The study duration has been revised; subjects will complete the study after 24 months of treatment with study drug.
- 18. The target blood Phe concentration has been revised from 480 μmol/L to 120-600 μmol/L for consistency with Study PAL-002.

- 19. The efficacy analysis has been revised to include assessment of subjects who maintain a target Phe concentration. Subjects to be included in the safety analysis population have been revised for clarity; subjects who have postdose safety information will be included in the safety analysis.
- 20. PK, blood Phe, and tyrosine assessments have been revised for subjects who are on a stable dosing regimen for at least 3 months; subjects may have these assessments performed less frequently (ie, at the monthly versus weekly visits).
- 21. The timing of the Early Termination visit has been revised from 1 week to 4 weeks after the final dose of study drug to allow for an assessment that was recommended by an allergy advisory board prior to study termination.
- 22. Collection of subject's allergy history has been added at the Screening visit.
- 23. A chest X-ray has been added to the 12-month and 24-month visits.
- 24. Information regarding an Interactive Voice Response System (IVRS) has been removed; study drug assignment will not be conducted using an IVRS.
- 25. The Medical Monitor has been changed.
- 26. The Schedule of Events and the Study Procedure section (Section 12.3) have been updated to reflect the changes to this amendment. In addition, assessment schedules have been added for subjects who increase their dose frequency to 2x/week and daily (Interim Dosing Visit).
- 27. Administrative revisions have been made to improve clarity and consistency.



**PAL-003** 


## PROTOCOL AMENDMENT TEXT REVISIONS

The following table summarizes the revisions made to the protocol and relates the changes to the appropriate rationale. Text that has been added or inserted is indicated by <u>underlined</u> font, and deleted text is indicated by <u>strikethrough</u> font.

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| Section 2/Synopsis<br>(Objectives) | The primary objective of the study is: • To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU. | | 1, 13, 27 |
| | The secondary objectives of the study are: • To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU who participated in Study PAL 002. | | |
| Section 2/Synopsis<br>(Study Design and Plan) | This is a long-term extension of a Phase 2, open-label, dose-finding study (Study PAL-002) in approximately 35-50 35 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002. | | 2, 13, 18, 27 |
| | Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety as determined by blood Phe concentrations. If a subject's blood Phe concentration is <120 µmol/L, the subject's diet may be adjusted to increase the amount of dietary Phe intake to maintain target blood Phe concentrations of 120-600 µmol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. | | |
| Section 2/Synopsis<br>(Study Design and Plan) | At least one interim analysis may be performed by the sponsor during the study. In addition to the Sponsor, aA Data Monitoring Committee (DMC) will monitor the study safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor. | | 11, 17, 18, 27 |
| | PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to | | |


**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | take rAvPAL-PEG. PAL-002 <u>subjects'</u> <u>participants'</u> rAvPAL-PEG dosing will continue in PAL-003 without interruption of <u>weekly</u> -dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations <u>of below 120-600480</u> µmol/L. <u>Subjects will continue to receive injections in the clinic, administered by clinic staff but may later be allowed to self administer doses of study drug at home. Whether a subject may be allowed to self administer study drug <u>dD</u>oses will be evaluated on an individual basis.</u> | | |
| | The dose may be modified at any time for safety. | | |
| | Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been controlled to within a target range (below 120-600480 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed but not to exceed 3x/week (fingerstick tests may be performed more frequently). | | |
| | A subject will continue in PAL-003 until one of the following occurs: | | |
| | 1. The subject withdraws consent and discontinues from the study. | | |
| | 2. The subject is discontinued from the study at the discretion of the Investigator. | | |
| | 3. The drug becomes commercially available following the appropriate marketing approval. The subject has completed the study through the Month 24 visit. | | |
| | 4. The study is terminated. | | |
| Section 2/Synopsis<br>(Study Design and Plan) | Dose Modifications: After any modifications (increases or decreases) to dose level or frequency, subjects should remain in the clinic for observation for at least 2 hours following the injection of study drug. The Investigator should remain at the site to assess the subject for safety. | | 2, 11, 27 |
| | Dose Adjustment-Increase Methodology: | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. <u>Decisions regarding dose increases will depend on available blood Phe and drug concentrations.</u> | | |
| | Blood Phe levels will be measured 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed. Subjects must have blood Phe concentration tested 3 days after a dose adjustment. There must be a minimum of 2 weeks after each dose adjustment before any additional dose adjustments may be made, so that blood Phe concentrations can be assessed. | | |
| | Depending upon the response to rAvPAL-PEG in PAL-002, an individual subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows. | | |
| | <ul> <li>The dose may be increased by increments of no more than 10-fold higher than<br/>the subject's current dose.</li> </ul> | | |
| | • When adjusting increasing the dose, a dose may be used that is between the dose cohort levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.3, 0.6, and 1.0 mg/kg) that were defined in the previous study (PAL-002). | | |
| | • The dose_may be adjusted by increasing the frequency up to daily-ofnumber of injections per week, up to one dose per day, for a maximum total weekly dose per week of not to exceed 2.0 mg/kg, including subjects who receive more than 1 dose/week. Subjects who have increased their dose frequency will have additional assessments performed (Interim Dosing Visit). | | |
| | • When a dose is <u>adjustedincreased</u> (either by <u>increasingehanging</u> the dose level or by <u>increasingehanging</u> the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time. | | |
| | • Only 1 dose adjustment is allowed every 2 weeks. | | |
| | • Blood Phe levels will be measured 3 days after each dose increase (fingerstick is | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | acceptable); more frequent or daily blood Phe measurements may be performed. | | |
| | <ul> <li>The dose may be decreased as appropriate to achieve or maintain a favorable<br/>blood Phe concentration for safety.</li> </ul> | | |
| | Dose Decrease Methodology | | |
| | A subject's diet should be assessed prior to any dose decreases. Changes to diet should only be made if blood Phe concentrations are <120 µmol/L. If a subject's blood Phe level is <120 µmol/L, the subject's dietary Phe intake should be increased to achieve a stable blood Phe concentration of 120-600 µmol/L. If the subject's blood Phe level is <120 µmol/L despite a high Phe diet, the rAvPAL-PEG dose will then be decreased. The subject will be asked about any changes to diet prior to any dose adjustments, and any changes to diet should be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. | | |
| | All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (>30% change from baseline) and drug concentrations, as well as toxicity (any hypersensitivity reaction). Dose decreases may occur for safety (ie, blood Phe concentration <120 $\mu$ mol/L) or other toxicity that may be improved with a lower, more frequent dose. | | |
| | A dose should first be reduced by dose level (1.0, 0.6, 0.3, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced. | | |
| Section 2/Synopsis<br>(Study Design and Plan | Stopping Criteria: If an individual subject exhibits drug related toxicity of a treatment-emergent CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. | | 6 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | The subject's data will be evaluated by the Principal Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level. | | |
| | In addition, if 2 or more subjects at a dose level exhibit drug related toxicity of a treatment-emergent CTCAE grade 3 or greater, further dosing of subjects at that dose level will be halted and no subjects will be treated at a any higher dose levels will be halted until a safety assessment is completed. In addition, the Food and Drug Administration (FDA) will be notified of this occurrence. | | |
| Section 2/Synopsis<br>(Number of Planned<br>Subjects) | 35 <u>-50</u> 35 subjects. | | 13, 27 |
| Section 2/Synopsis<br>(Diagnosis and All<br>Criteria for Inclusion and<br>Exclusion) | Numbering has been added to all of the criteria. | | 27 |
| Section 2/Synopsis<br>(Diagnosis and All | Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study: | | 27 |
| Criteria for Inclusion and Exclusion) | 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation. | | |
| | 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL 001 or PAL-002. | | |
| Section 2/Synopsis | rAvPAL-PEG doses will be administered SC and the favorable dose (the dosage that provides control of blood Phe concentrations within the target range of 120-600 µmol/L | | 18, 27 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| (Investigational Product,<br>Dose, Route and<br>Regimen) | for a minimum of 2 weeks) will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. | | |
| Section 2/Synopsis (Duration of Treatment) | 3. The drug becomes commercially available following the appropriate marketing approval. The subject has completed the study through the Month 24 visit. | | 17 |
| Section 2/Synopsis<br>(Criteria for Evaluation) | Immunogenicity: The presence of antibodies will be assessed. | | 27 |
| Section 2/Synopsis<br>(Safety Analysis) | All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses. | | 19 |
| Section 2/Synopsis<br>(Efficacy Analysis) | Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 120-600 µmol/L will be summarized by each scheduled time point. | | 19 |
| Section 2/Synopsis<br>(Pharmacokinetic<br>Analysis) | Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 120-600480 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks. Should data become available from PAL-002 that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed but not to exceed 3x/week. | | 3, 18 |
| Section 2.1/Schedule of Events (Table 2.1: | The Schedule of Events has been revised to reflect changes to the study procedures. The Final F/U and Early Termination visits have been separated, and | | 8, 10, 15, 20,<br>21, 22, 23, 26 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Schedule of Events) | an Unscheduled Hypersensitivity Reaction Visit has also been added. | | |
| | Tables 2.1.2 (Interim Dosing Visit Schedule, Subjects Whose Dose Is Increased to 2x/Week) and 2.1.3 (Interim Dosing Visit Schedule, Subjects Whose Dose Is Increased to Daily) have been added. | | |
| Section 4/List of | CBC complete blood count | | 27 |
| Abbreviations and Definition of Terms | CH50 total hemolytic complement | | |
| | <u>C<sub>max</sub></u> maximum plasma concentration | | |
| | <u>CRP</u> <u>C-reactive protein</u> | | |
| | CTCAE Common Terminoallogy Criteria for Adverse Events | | |
| | C <sub>trough</sub> predose concentration of rAvPAL PEG | | |
| | DCF Data Clarification Form | | |
| | IND Investigational New Drug | | |
| | IVRS interactive voice response system | | |
| | IgE immunoglobulin E | | |
| | NOAEL no observable adverse effect level | | |
| | rAvPAL-PEG <u>rAv</u> phenylalanine ammonia lyase <u>-PEG</u> | | |
| Section 6/Investigators | The study will be administered by and monitored by employees or representatives | | 27 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| and Study Administrative | of BioMarin. Clinical Research Associates (CRAs) or trained designees will | | |
| Structure | monitor each site on a periodic basis and perform verification of source | | |
| | documentation for each subject as well as other required review processes. | | |
| | BioMarin's Regulatory Affairs Department (or designee) will be responsible for | | |
| | the timely reporting of serious adverse events (SAEs) to appropriate regulatory | | |
| | authorities as required. Some study assessments, including administration of study | | |
| | drug, may be performed at the subject's home. All assessments performed for this | | |
| | study will be administered by clinic staff or other qualified and trained study | | |
| | personnel. | | |
| Section 7.1/Nonclinical<br>Studies | Weekly subcutaneous (SC) administration of 80 mg/kg of rAvPAL-PEG (approximately 4 IU/mouse) for greater than 2 to 3 months lowered and stabilized plasma blood-Phe concentration from approximately 2000 μM to less than 200 μM. | | 5, 27 |
| | The safety of rAvPAL-PEG was evaluated in safety pharmacology studies (respiratory, central nervous system [CNS] and cardiovascular [CV]) and toxicity with toxicokinetic studies (single and 28-day repeated dose) in rats and cynomolgus monkeys. Overall, in the nonclinical in all toxicity studies, no immune related toxicities anaphylactoid-like reactions or injection-site reactions | | |
| | were noted were seen either systemically or at the injection site. No specific polyethylene glycol (PEG)-related histological findings were observed during the 28-day repeated dose studies. | | |
| | The main finding in the 28-day study was the possible drug-related observation of | | |
| | minimal to slight degeneration of blood vessels of predominantly medium-sized | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | muscular arteries with a non-dose-dependent involvement of different organs | | |
| | observed in 1 male in the 0.1 mg/kg and 1 male and 1 female in the 1.0 mg/kg | | |
| | rAvPAL-PEG dose groups. No degeneration of the arteries was observed in either | | |
| | the control or animals administered 0 and 0.01 mg/kg rAvPAL-PEG. | | |
| Section 7.1/Nonclinical | Chronic repeat-dose toxicity and toxicokinetic studies were conducted in the rat | | 5 |
| Studies | (17/26 weeks) and monkey (39 weeks). In the 26-week study of rats, weight loss | | |
| | was observed in the rats given 25 mg/kg/dose of rAvPAL-PEG, SC; | | |
| | corresponding decreased food consumption was observed in the males. The main | | |
| | histological finding was focal-to-multifocal areas of vacuolar degeneration of | | |
| | renal tubule cells in the kidney of 3 males given 25 mg/kg and 3 females given | | |
| | ≥8 mg/kg rAvPAL-PEG. This renal tubule finding persisted in the kidney of both | | |
| | sexes given $\geq 8$ mg/kg/dose at the end of the 12-week recovery phase without | | |
| | evidence of reversibility. Increased vacuolation was observed in histiocytic cells | | |
| | of the liver, spleen, mesenteric lymph node, mandibular lymph node, and adrenal | | |
| | cortex of males given 25 mg/kg/dose and females given ≥8 mg/kg/dose; | | |
| | vacuolation of histiocytic cells in the testes were also observed in males given | | |
| | 25 mg/kg/dose. Both renal tubule vacuolation and histiocytic cell vacuoles have | | |
| | been associated with PEG-related catabolism and administration of other | | |
| | PEGylated proteins. | | |
| | In the 39-week, chronic repeat-dose toxicity and toxicokinetic study in monkeys, | | |
| | dose levels of 7.0 and 5.0 mg/kg/dose rAvPAL-PEG were not tolerated in female | | |
| | monkeys and resulted in body weight loss, decreased food consumption, and | | |

**PAL-003** 


| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | hypoactivity. The only adverse microscopic finding was arterial inflammation of | | |
| | small and mid-sized arteries in multiple organs and/or tissues in most animals that | | |
| | were given ≥3 mg/kg/dose rAvPAL-PEG SC twice weekly at the end of the | | |
| | dosing phase. The inter-individual organ involvement was highly variable; some | | |
| | animals had findings in one organ and others had multiple organs with arterial | | |
| | inflammation. Additionally, not all arteries had signs of inflammation and arterial | | |
| | inflammation was resolved by the end of the 13-week recovery period. A full | | |
| | analysis of these findings including the involvement of the anti-drug antibodies, | | |
| | antibody isotypes, PEG distribution, and rAvPAL-PEG is ongoing. The no | | |
| | observable adverse effect level (NOAEL) for the 17-week and 39-week studies, in | | |
| | rat and monkey, respectively, is 1 mg/kg/dose. The NOAEL from these studies | | |
| | represents greater than a 100-fold safety factor over the starting dose in PAL-002. | | |
| Section 7.2/Previous | This study is an extension of the second human clinical study with rAvPAL-PEG | | 27 |
| Clinical Studies | (Study PAL-002). Study PAL-001, the first-in-human clinical study of | | |
| | rAvPAL-PEG, was designed as a Phase 1, open-label, single-dose, | | |
| | dose-escalation study in approximately 3525 subjects, 16 to 50 years old, with | | |
| | PKU. The doses for this study are <u>based on data from nonclinical studies and</u> | | |
| | PAL-001 and are planned to be in the same range as those tested in PAL-001 and | | |
| | PAL 002 (0.001 through 1.0 mg/kg per injection (not to exceed 2.0 mg/kg/week), | | |
| | provided no dose-limiting toxicity was observed in those studies Study PAL-002. | | |
| Section 7.4/Summary of | It is not expected that data from PAL 001 and PAL-002 will change the | | 4, 27 |
| Overall Risks and Benefits | assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant | | |


**PAL-003** 

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | PEGylated non-human enzymes currently in use. | | |
| Section 7.4.1/Toxicity Due to Exposure to PEG | No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg of SC rAvPAL-PEG SC. | | 27 |
| Section 7.4.2/Toxicity Due to an Immunologic Reaction | This section has been reorganized to include updated safety information from Study PAL-001. Presentation of information in this section, including section numbers, has also been revised. | | 27 |
| Section 7.4.2/Toxicity Due to an Immunologic Reaction | The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. In animal models, the immune response against the foreign protein PAL in rAvPAL PEG has been mitigated by PEGylation. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). Administration of rAvPAL-PEG may lead to anti-PEG antibody formation, and the duration of this possible effect is not known. This may limit a subject's future ability to be treated with other PEG-containing (eg, Depo-Provera) or PEGylated (eg, PEG-interferon) injectable drugs. It is therefore recommended that any PEG-containing injectable drug administered to subjects after completion of this study be done under medical observation. | | 4, 27 |
| Section 7.4.2.1/ Reactions with Depo ProveraSystemic Skin Reactions | Two subjects enrolled in PAL 001 who had received one dose of rAvPAL PEG experienced hypersensitivity reactions to intramuscular (IM) Depo Provera, a contraceptive containing PEG 3350. Both subjects had previously received multiple IM Depo Provera injections without complications. The first subject, a year old developed bruising at the injection site on Day 1 that resolved on Day 15. | | 4, 27 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | difficulty 10 minutes after receiving IM Depo-Provera given 40 days after | | |
| | rAvPAL PEG injectionwas treated in the emergency room with | | |
| | the events the state of the sta | | |
| | resolved the same day, and the subject had no further complications. The subject | | |
| | had no prior history of any reactions to Depo Provera. Subsequently, while under | | |
| | the care of an allergist/immunologist, the subject had a mild reaction to a | | |
| | concentrated intradermal (1:10) exposure of Depo Provera. was later given a | | |
| | full dose of IM Depo Provera without problems. | | |
| | The second subject, an year old , had a slightly raised, erythematic rash | | |
| | below the site of rAvPAL PEG injection on Day 11 that resolved without | | |
| | treatment on Day 15. developed generalized hives on arms and legs and | | |
| | mild difficulty breathing 20 minutes after receiving IM Depo Provera (and | | |
| | third dose of Gardasil) given 15 days after rAvPAL-PEG injection. | | |
| | symptoms subsided after received oral given by mother. | | |
| | not visit the emergency room. The subject had no prior history of any reactions to | | |
| | Depo Provera or Gardasil (Gardasil dose not contain PEG). was subsequently | | |
| | seen by an allergist/immunologist, and the results are pending. | | |
| | Because Depo Provera contains PEG 3350 as an excipient, it is possible that the | | |
| | administration of rAvPAL PEG caused anti PEG antibody formation that led to a | | |
| | cross reaction with Depo Provera in these subjects. Therefore, it is possible that | | |
| | prior exposure to rAvPAL PEG might sensitize subjects to other PEG containing | | |
| | injectable drugs. Alternatively, the presence of Depo Provera could have led to | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | antibody formation and cross-reaction with rAvPAL-PEG, leading to rAvPAL- | | |
| | PEG injection site reactions. Since it is currently unknown whether Depo Provera | | |
| | has a sensitizing effect to PEG and the exact basis for these reported events is not | | |
| | known, the use of PEG containing injectable drugs prior to and during the study is | | |
| | prohibited as a precautionary measure (refer to the addendum and Sections 9.3.2 and 9.4.8). | | |
| | Two subjects who were enrolled in Study PAL-001 and received the | | |
| | protocol-defined single dose of rAvPAL-PEG reported systemic skin reactions | | |
| | (generalized skin rash) that were attributed to treatment with study drug. One | | |
| | subject received a single dose of 0.001 mg/kg rAvPAL-PEG, and the other subject | | |
| | received a single dose of 0.01 mg/kg rAvPAL-PEG. Both of these events were | | |
| | reported as serious and followed administration of Depo-Provera injections | | |
| | (medroxyprogesterone injection), an injectable contraception. These allergic | | |
| | reactions are thought to be related to the PEG molecules that are found in both the | | |
| | study drug, rAvPAL-PEG, and Depo-Provera. These reactions are not likely to be | | |
| | experienced concurrent with other birth control medications. | | |
| | The 2 subjects were administered study drug during PAL-001 and then | | |
| | experienced an allergic reaction following an injection of Depo-Provera. The | | |
| | symptoms of the reactions were hives on the arms and legs and difficulty | | |
| | breathing. The symptoms for both subjects resolved within 1 day following | | |
| | treatment with medication, including the | | |
| | . Both subjects were examined by an allergy specialist after | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | they completed participation in PAL-001. A skin prick test with Depo-Provera | | |
| | was administered as part of this examination. One subject had a mild allergic | | |
| | reaction to the test; however, no further reactions or complications were reported | | |
| | following subsequent administration of a full dose of Depo-Provera. The subject | | |
| | continues to receive regular doses (every 3 months) of Depo-Provera, and no | | |
| | further reactions have been reported to date (15OCT2009). The second subject | | |
| | also had a positive reaction to Depo-Provera following administration of the skin | | |
| | prick test. When a subsequent full dose of Depo-Provera was administered, | | |
| | developed hives, itching, and chills. The subject's symptoms resolved within | | |
| | 1 day of taking medication prescribed by an allergist. | | |
| | The active drug substance in rAvPAL-PEG is a bacterial protein that may elicit | | |
| | immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and | | |
| | others. It is possible that the physio-chemical properties of rAvPAL-PEG may | | |
| | induce immunologic sensitization to the protein rAvPAL and to PEG. Although | | |
| | results from nonclincal studies of rAvPAL-PEG conducted in rats and | | |
| | cynomolgus monkeys did not indicate signs of immune-mediated toxicities, it is | | |
| | possible that the physio-chemical properties of rAvPAL-PEG may induce | | |
| | immunologic sensitization to the protein rAvPAL and to PEG in humans. Since iIt | | |
| | is currently unknown whether administration of PEG-containing drugs, such as | | |
| | Depo-Provera, has a sensitizing effect to PEG in rAvPAL-PEG when | | |
| | administered in humans. Because and the exact basis for these reported events and | | |
| | their duration is not known, the use of PEG-containing injectable drugs prior to, | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | and during, and after this study is prohibited as a precautionary measure (refer to Sections 9.3.2 and 9.4.8.). | | |
| Section 7.4.2.2/<br>Management of Allergic<br>Reactions | Information regarding the management of local skin, large local skin, and systemic reactions is provided in Section 9.1.1. Detailed instructions for the management of allergic reactions are provided in the Study Reference Manual. | | 27 |
| Section 7.4.3/Effects of Low Blood Phe | If a subject's blood Phe concentration is too low, the subject's diet, current dose of study drug, or both may be adjusted. | | 1, 27 |
| Section 8/Study<br>Objectives | To evaluate the effect of long-term administration of <u>multiple doses of SC</u> injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU. | | 1, 13, 27 |
| | The secondary objectives of the study are: • To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU who participated in Study PAL 002. | | |
| Section 9.1/Overall Study<br>Design and Plan | This is a long-term extension of a Phase 2, open-label, dose-finding study (PAL-002) in approximately 35-50 35 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002. | | 2, 13, 27 |
| | Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety as determined by blood Phe concentrations. If a subject's blood Phe | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | concentration is <120 µmol/L, the subject's diet may be adjusted to increase the | | |
| | amount of dietary Phe intake to maintain target blood Phe concentrations of | | |
| | 120-600 μmol/L. Changes to diet will be made per the discretion of the Investigator | | |
| | in consultation with the Sponsor's Medical Officer. For information regarding | | |
| | changes to diet for safety and decreases in dose, refer to Section 9.1.2.2. | | |
| Section 9.1/Overall Study | At least one interim analysis may be performed by the sponsor during the study. | | 11, 17, 18, 27 |
| Design and Plan | In addition to the Sponsor, aA Data Monitoring Committee (DMC) will monitor | | |
| | the study safety of subjects in the study. The DMC is an independent committee | | |
| | that will act in an advisory capacity to the Sponsor. | | |
| | PAL-003 is designed to evaluate long-term treatment of subjects who are | | |
| | continuing to take rAvPAL-PEG. PAL-002 subjects' participants' rAvPAL-PEG | | |
| | dosing will continue in PAL-003 without interruption of weekly dosing. In PAL- | | |
| | 003, each subject's dose will be adjusted as needed to attain or maintain blood | | |
| | Phe concentrations below of 120-600480 µmol/L based upon recommendations | | |
| | by the German Working Group for Metabolic Diseases (Burgard, 1999, Eur J | | |
| | Pediatr). Subjects will continue to receive injections in the clinic, administered by | | |
| | clinic staff., but may later be allowed to self administer doses of study drug at | | |
| | home. Whether a subject may be allowed to self administer study drug dDoses | | |
| | will be evaluated on an individual basis. All of the following criteria must be met | | |
| | before a subject may self administer doses of the study drug: | | |
| | The subject is willing and able to administer the study drug as directed. | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | The sponsor agrees that self-administration is appropriate. | | |
| | The subject has achieved a favorable dose (ie, the dosage that provides control of blood Phe concentrations within the target range for a minimum of 2 weeks). | | |
| | The dose may be modified at any time for safety. | | |
| | Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been controlled to within a target range (below 120-600480 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed but not to exceed 3x/week (fingerstick tests may be performed more frequently). A subject will continue in PAL-003 until one of the following occurs: 1. The subject withdraws consent and discontinues from the study. 2. The subject is discontinued from the study at the discretion of the Investigator. | | |
| | <ul> <li>3. The drug becomes commercially available following the appropriate marketing approval. The subject has completed the study through the Month 24 visit.</li> <li>4. The study is terminated.</li> </ul> | | |
| Section 9.1.1/ Management of Local and Systemic Reactions to rAvPAL-PEG | Presentation of information in this section, including section numbers, has been revised. | | 27 |
| Section | 9.1.1.1 Subjects Who Have <u>Had Experienced Previous Hypersensitivity</u> | | 7-9 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| 9.1.1/Management of | Reactions to rAvPAL-PEG or a PEG-Containing Product | | |
| Local and Systemic<br>Reactions to<br>rAvPAL-PEG | Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from PAL 001 or | | |
| | PAL-002 are excluded from participation in this study. Subjects who experienced | | |
| | a generalized skin rash are included in this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in PAL-002 are eligible to | | |
| | participate in this study. However, sSubjects may develop such systemic, large | | |
| | local skin, or local skin reactions after enrollment in PAL-003. Management of | | |
| | such reactions described below. Refer to Figure 9 1.1.2.2.1 for a flowchart for | | |
| | managing these subjects. Refer to Section 9.1.1.2 for definitions of local skin, | | |
| | large local skin, and systemic skin reactions. For management of hypersensitivity | | |
| | reactions that occur during this study, refer to Section 9.1.1.3 and | | |
| | Figure 9.1.1.3.1. | | |
| | 9.1.1.2 Definition of Hypersensitivity Reactions to rAvPAL-PEG Administered Subcutaneously | | |
| | During Study PAL-003, subjects may experience hypersensitivity reactions to rAvPAL-PEG. The hypersensitivity reactions are defined as follows: Local skin reaction: | | |
| | • Skin signs or symptoms in 1 affected primary location, 1 affected location ie, hives, wheals, or swelling or an area of erythema, or redness, induration, pain, or itching at or near the site of injection. | | |

PAL-003

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | <ul> <li>Skin signs or symptoms, ie, hives, wheals, or swelling or an area of erythema, redness, or induration with pain or itching that extends beyond the site of injection by approximately 6 inches (15 cm) and/or signs or symptoms that are not contiguous to the injection site. These may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure and, therefore, will be managed as a systemic reaction when not contiguous to the injection site.</li> <li>Systemic reaction (including generalized skin symptoms):</li> <li>Skin and non-skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema, or anaphylaxis or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological.</li> <li>For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.</li> </ul> | | |
| | | | 7-9, 27 |



**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| 9.1.1.3.1/Local Skin | After enrollment in PAL 003, sSubjects who have had a local skin reaction (refer | | 7-9 |
| Reactions | to Section 9.1.1.2 for definition) after administration ofto rAvPAL-PEG in | | |
| | PAL-001, PAL-002, or this study or a PEG containing product willmay be | | |
| | premedicated orally with acetaminophen and antihistamines and/or oral steroids, | | |
| | 1 hour prior to study drug dosing. Recommended premedications are | | |
| | acetaminophen and antihistamine (Claritin-Zyrtec [cetirizine] is preferred). | | |
| | The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg Claritin | | |
| | Zyrtec or 25 to 50 mg Benadryl [diphenahydramine]; an example for steroids | | |
| | would be 70 mg oral prednisone). Because Benadryl can cause drowsiness, it may | | |
| | be administered only if the subject is accompanied by a designated driver. | | |
| | Symptoms of local reactions may be treated with local application of ice and | | |
| | non-sedating oral and/or topical antihistamines and/or topical steroids (refer to | | |
| | Section 7.4.2.2). | | |
| | If the local skin reaction worsens with a repeat injection (as determined by the | | |
| | Investigator in consultation with the Study Medical Officer) even with | | |
| | premedication prior to study drug dosing, the subject must be withdrawn from the | | |
| | study and complete an Early Termination Visit. | | |
| | 9.1.1.3.2 <u>Large Local Skin Reactions</u> | | |
| | If a subject has a local skin reaction, a digital photograph of the reaction should be | | |



**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | taken if possible. Large local skin reactions (refer to Section 9.1.1.2 for a | | |
| | definition) may or may not be contiguous to the rAvPAL-PEG injection site. | | |
| | The location of the large local skin reaction relative to the rAvPAL-PEG injection | | |
| | site will determine if a subject may remain in the study and continue to be | | |
| | administered rAvPAL-PEG. An example of a large local reaction that is not | | |
| | contiguous to the injection site is if an injection took place in the right upper arm | | |
| | and there are lesions beyond the elbow joint in the right forearm or lesions beyond | | |
| | the shoulder joint on the right trunk. | | |
| | Subjects who have large local skin reactions that are contiguous to the injection | | |
| | site may remain in the study. Subjects who have large local skin reactions that are | | |
| | not contiguous to the injection site may have additional assessments performed | | |
| | (Unscheduled Hypersensitivity Reaction Visit) per Investigator discretion and | | |
| | must then be terminated from the study. A decision to terminate a subject from | | |
| | the study must be agreed to by both the Investigator and the Sponsor's Medical | | |
| | Officer. | | |
| | 9.1.1.3.2.1 <u>Large Local Skin Reactions Contiguous to Injection Site</u> | | |
| | Subjects who develop a large local skin reaction contiguous to the injection site | | |
| | after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing | | |
| | product may remain in the study. Large local skin reactions that are contiguous to | | |
| | the injection site should be managed as local skin reactions (refer to | | |
| | Section 9.1.1.3.1). For the remainder of the study, subjects must be premedicated | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | orally with acetaminophen and antihistamines 1 hour prior to study drug dosing. | | |
| | Recommended premedications are acetaminophen and antihistamine (Zyrtec | | |
| | [cetirizine] is preferred). The dosage will be standard (eg, 1000 mg | | |
| | acetaminophen and 10 mg Zyrtec or 25 to 50 mg Benadryl [diphenahydramine]). | | |
| | Because Benadryl can cause drowsiness, it may be administered only if the | | |
| | subject is accompanied by a designated driver. | | |
| | Symptoms of large local skin reactions may be treated with local application of | | |
| | ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to | | |
| | Section 7.4.2.2). | | |
| | 9.1.1.3.2.2 <u>Large Local Skin Reactions Not Contiguous to Injection Site</u> | | |
| | Large local skin reactions that are not contiguous to the injection site may be | | |
| | associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure | | |
| | to rAvPAL-PEG and, therefore, will be managed as a systemic reaction. Subjects | | |
| | who develop large local skin reactions that are not contiguous to the injection site | | |
| | after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing | | |
| | product may not continue to participate in the study. Subjects may have additional | | |
| | assessments performed (ie, Unscheduled Hypersensitivity Skin Reaction Visit) | | |
| | immediately after the reaction (within 48 hours): serum anti-rAvPAL-PEG | | |
| | antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL immunoglobulin M | | |
| | [IgM], anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, | | |
| | and anti-rAvPAL-PEG immunoglobulin E [IgE]); serum tryptase level; | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Section 100/1100 | sedimentation rate; C-reactive protein (CRP), total hemolytic complement | Comments | Change 140. |
| | (CH50), and complements $C_1$ and $C_4$ ; and clinical laboratory tests (urinalysis, | | |
| | chemistry, hematology). Subjects will then be terminated from the study and | | |
| | should be scheduled to complete the Early Termination Visit (refer to | | |
| | Section 12.4). | | |
| | Symptoms of large local skin reactions may be treated with local application of | | |
| | ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to | | |
| | Section 7.4.2.2). | | |
| Section 9.1.1.3.3/ | After enrollment in PAL 003, subjects who have a systemic reaction that includes | | 7, 8, 27 |
| Systemic Reactions | noncutaneous systemic symptoms, such as respiratory problems, hypotension, or | | |
| | angioedema, to rAvPAL PEG or a PEG containing product will be evaluated with | | |
| | a skin prick test. If the test is positive, the subject will be excluded from the study. | | |
| | Subjects with prior systemic reactions that included only skin manifestations to | | |
| | rAvPAL PEG or a PEG containing product after PAL 003 enrollment will be | | |
| | premedicated with acetaminophen and antihistamines and/or oral steroids (one | | |
| | hour prior to study drug dosing) and will continue to receive rAvPAL PEG. | | |
| | Reactions to skin prick testing or rAvPAL PEG administered SC are defined as follows: | | |
| | Local reaction: 1 affected location, ie, hives, wheals, or swelling or an area of | | |
| | erythema or redness at or near the site of injection. | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | Systemic reaction: more than 1 affected location, ie, cutaneous reaction in more | | |
| | than 1 area, and/or any other generalized symptoms, such as hypotension, | | |
| | angioedema or anaphylaxis or the involvement of other organ systems (eg, | | |
| | respiratory, cardiovascular, gastrointestinal). | | |
| | Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a | | |
| | definition) after administration of rAvPAL-PEG will be terminated from the | | |
| | study. Subjects who experience generalized skin symptoms are included in this | | |
| | category. Immediately after the systemic reaction (within 48 hours), subjects with | | |
| | generalized skin symptoms must have additional assessments performed for | | |
| | safety (ie, Unscheduled Hypersensitivity Skin Reaction Visit): serum | | |
| | anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, | | |
| | anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG | | |
| | IgE); serum tryptase level (optional; it is recommended that this sample be drawn | | |
| | immediately after reaction); sedimentation rate; CRP, CH50, C <sub>1</sub> , and C <sub>4</sub> ; and | | |
| | clinical laboratory tests (urinalysis, chemistry, hematology; refer to | | |
| | Figure 9.1.1.3.1). Subjects who have a systemic reaction without generalized skin | | |
| | symptoms may have these assessments performed per Investigator discretion. | | |
| | Subjects will then be terminated from the study and should be scheduled to | | |
| | complete the Early Termination Visit (refer to Section 12.4). | | |
| Section 9.1.2/Dose | After any modifications (increases or decreases) to dose level or frequency, | | 2, 27 |
| Modifications | subjects should remain in the clinic for observation for at least 2 hours following | | |
| | the injection of study drug. The Investigator should remain at the site to assess the | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | subject for safety. | | |
| Section 9.1.2.1/Dose<br>Increase Methodology | Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. <u>Decisions regarding dose increases</u> will depend on available blood Phe and drug concentrations. | | 2, 11, 27 |
| | Depending upon the response to rAvPAL-PEG in PAL-002, <u>an individual</u> subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows: | | |
| | • The dose may be increased by increments of no more than 10-fold higher than the subject's current dose. | | |
| | • When adjusting increasing the dose, a dose may be used that is between the dose eohort levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.3, 0.6, and 1.0 mg/kg) that were defined in the previous study (PAL-002). | | |
| | • The dose may be adjusted by increasing the frequency up to daily of number of injections per week, up to one dose per day, for a maximum total weekly dose per week of not to exceed 2.0 mg/kg, including subjects who receive more than 1 dose/week. Subjects who increase their dose frequency should perform the Interim Dosing Visit assessments (refer to Section 12.3.5 and Tables 2.1.2 and 2.1.3). | | |
| | • When a dose is <u>adjustedincreased</u> (either by <u>increasingehanging</u> the dose level or by <u>increasingehanging</u> the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time. | | |
| | • Only 1 dose adjustment is allowed every 2 weeks. | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | Blood Phe levels will be measured 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed. | | |
| | The dose may be decreased as appropriate to achieve or maintain a favorable blood Phe concentration for safety. | | |
| | Subjects must have blood Phe concentration tested 3 days after a dose adjustment. | | |
| | There must be a minimum of 2 weeks after each dose adjustment before any | | |
| | additional dose adjustments may be made, so that blood Phe concentrations can | | |
| | be assessed. | | |
| | 9.1.2.2 <u>Dose Decrease Methodology</u> | | |
| | A subject's diet should be assessed prior to any dose decreases. Changes to diet | | |
| | should only be made if blood Phe concentrations are <120 μmol/L. If a subject's | | |
| | blood Phe level is <120 μmol/L, the subject's dietary Phe intake should be | | |
| | increased to achieve a stable blood Phe concentration of 120-600 μmol/L. If the | | |
| | subject's blood Phe level is <120 μmol/L despite a high Phe diet, the | | |
| | rAvPAL-PEG dose will then be decreased. The subject will be asked about any | | |
| | changes to diet prior to any dose adjustments, and any changes to diet should be | | |
| | made per the discretion of the Investigator in consultation with the Sponsor's | | |
| | Medical Officer. | | |
| | All dose decreases must be agreed to by both the Investigator and the Sponsor's | | |
| | Medical Officer. Decisions regarding dose decreases will depend on available | | |
| | information regarding a subject's blood Phe (>30% change from baseline) and | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | drug concentrations, as well as toxicity (any hypersensitivity reaction as defined | | |
| | in Section 9.1.1.2). Dose decreases may occur for safety (ie, blood Phe | | |
| | concentration < 120 μmol/L) or other toxicity that may be improved with a lower, | | |
| | more frequent dose. | | |
| | A dose should first be reduced by dose level (1.0, 0.6, 0.3, 0.1, 0.06, 0.03, 0.01, | | |
| | 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these | | |
| | specified dose levels. If further dosing adjustments are required to attain the target | | |
| | Phe concentration, dosing frequency may be reduced. | | |
| Section 9.1.3/Stopping | If an individual subject exhibits drug related toxicity of a treatment-emergent | | 6 |
| Criteria | CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity | | |
| | resolves. The subject's data will be evaluated by the Principle Investigator (PI) | | |
| | and the Study Medical Officer, and a decision will then be made whether to | | |
| | discontinue the subject from the study, restart dosing at the same dose level, or | | |
| | restart dosing at a lower dose level. | | |
| | In addition, if 2 or more subjects at a dose level exhibit <del>drug related</del> toxicity of <u>a</u> | | |
| | treatment-emergent CTCAE grade 3 or greater, further dosing of subjects at that | | |
| | dose level will be halted and no subject will be treated at a any higher dose levels | | |
| | will be halted until a safety assessment is completed. In addition, the Food and | | |
| | Drug Administration (FDA) will be notified of this occurrence. | | |
| Section 9.3.2/Exclusion | 3. Use or planned use of any injectable drugs containing PEG (other than | | 27 |
| Criteria | rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | during study participation. | | |
| | 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including | | |
| | hypersensitivity reactions that necessitated early termination from PAL-002. | | |
| Section 9.3.4/Subject | After enrollment of 35 subjects, if any single cohort (identified during PAL 002) | | 13, 27 |
| Identification and | has less than 3 subjects due to early terminations, those subjects will be replaced. | | |
| Replacement of Subjects | Replacement subjects will enter the study at the same dose cohort level as the | | |
| | subject they are replacing. | | |
| | Each subject was assigned a unique subject identifier in either PAL 001 or | | |
| | PAL 002. Subjects will retain the same subject number <u>assigned</u> used in | | |
| | PAL-002. This unique identifier will be on all case report form (CRF) pages. In | | |
| | legal jurisdictions where use of initials is not permitted, a substitute identifier will | | |
| | be used. | | |
| | Subjects who do not complete the study will not be replaced. | | |
| | This unique identifier will be on all case report form (CRF) pages. In legal | | |
| | jurisdictions where use of initials is not permitted, a substitute identifier will be | | |
| | used. | | |
| Section 9.4.4/Directions | Study drug will be administered by clinic staff or other qualified and trained study | | 11, 27 |
| for Administration | personnel. | | |
| | Table 9.4.4.1 Number of Injections Required For an Individual | | |
| | Weighing 80 kg | | |



**PAL-003** 

| Section No./Title | Revision | | | | Comments | Relates to Change No. |
|---|---|---|---|---|---|---|
| | Dose Group<br>(mg/kg) | Weight (kg) | Volume of Study Drug (mL) <sup>a</sup> | No. of<br>Injections <sup>b</sup> | | |
| | 0.001 | 80 | 0.8 | 1 | | |
| | 0.003 | 80 | 0.6 | 1 | | |
| | 0.01 | 80 | 0.8 | 1 | | |
| | 0.03 | 80 | 0.2 | 1 | | |
| | 0.06 | <u>80</u> | 0.5 | <u>1</u> | | |
| | 0.1 | 80 | 0.8 | 1 | | |
| | 0.3 | 80 | 2.4 | 2 | | |
| | 0.6 | <u>80</u> | 4.8 | <u>2 or 3</u> | | |
| | 1.0 | 80 | 8.0 | 4 | | |
| | The state of the s | | nere to the study drug admini | | | |
| | • | | eduled doses of study drug, l | ooth dose level and | : | |
| | dose frequency will | l need to be re- | evaluated. | | | |
| Section 9.4.5/Method of<br>Assigning Subjects to<br>Treatment Groups | An interactive voice assigned dose and s | | em (IVRS) will be used to transfer. | ek subjects' | | 24 |
| Section 9.4.6/Selection of | This Phase 2 study | aims to evaluat | e the efficacy, safety, tolerab | ility, and PK | | 18, 27 |
| Doses Used in the Study | * | • | vPAL-PEG after long-term a | | | |
| | | | ose that produces a reduction | | | |
| | concentrations to be | <del>elow</del> 120-60048 | 80 μmol/L will be determined | I for each subject. | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | The doses for this study are based upon the results of nonclinical studies and | | |
| | PAL-001. Findings in cynomolgus monkeys dosed with a single administration of | | |
| | 60 mg/kg rAvPAL PEG included severe morbidity, decreased plasma Phe | | |
| | concentration, decreased protein synthesis, and GI lesions. Plasma Phe | | |
| | concentrations were reduced to below the level of detection in the lower dose | | |
| | groups, without other findings (refer to Section 7.1). The no observable adverse | | |
| | effect level (NOAELs) from nonclinical studies in rats and monkeys represents a | | |
| | greater than 100-fold safety factor over the starting dose administered in PAL- | | |
| | 002, (0.001 mg/kg). The doses for this study will be based upon the results of | | |
| | PAL 001 and PAL 002. | | |
| Section 9.4.6.1/Selection | Study drug will be administered in the morning by clinic staff or other qualified | | 11, 27 |
| of Timing of Dose for<br>Each Subject | and trained study personnel or by the subject, if appropriate. | | |
| Section 9.4.8/Prior and | Use or planned use of any injectable drugs containing PEG (other than | | 7-9, 27 |
| Concomitant Medications | rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to | | |
| | Screening and during study participation. A list of PEG-containing injectable | | |
| | drugs is provided in the study reference materials. Subjects who have had a prior | | |
| | local skin reaction to rAvPAL-PEG or a PEG-containing product will be | | |
| | premedicated with acetaminophen and antihistamines and/or oral steroids (refer to | | |
| | Section 9.1.1). If the local skin reaction worsens with a repeat injection (as | | |
| | determined by the Investigator in consultation with the Study Medical Officer) | | |
| | even with premedication prior to study drug dosing, the subject must be | | |


| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | withdrawn from the study and complete an Early Termination Visit. Subjects who have had a prior systemic hypersensitivity reaction to rAvPAL-PEG or a PEG-containing product are excluded from participation in this study will be premedicated with acetaminophen and antihistamines and/or oral steroids (refer to Section 9.1.1). If the local or systemic reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study. | | |
| Section 9.6/Dietary or<br>Other Protocol<br>Restrictions | Subjects will be instructed that diet should not be altered during the course of the study except as necessary for safety. If a subject's blood Phe concentration is <120 µmol/L, the subject's diet will be adjusted to maintain blood Phe concentrations of 120-600 µmol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next dose of study drug. The dietary record will be maintained with the study source documents. | | 2, 15, 27 |

**PAL-003** 

| Section No./Title | Revision | | | Comments | Relates to Change No. |
|---|---|---|---|---|---|
| Section 9.7.1/Efficacy | <b>Table 9.7.1.1: Sun</b> | nmary of Laboratory As | sessments | | 27 |
| and Safety Measurements Assessed | Laboratory Assessment | Party Responsible for Performing Test | Section in<br>Protocol for<br>Details | | |
| | Clinical laboratory tests | Central laboratory | 9.7.5 | | |
| | Antibody testing | BioMarin <sup>a</sup> | 9.7.4.2 | | |
| | PK variables | <del>Central</del><br><del>laboratory</del> BioMarin | 9.7.3 | | |
| | Blood Phe concentrations | Central laboratory | 9.7.2.1 | | |
| | Urinalysis, pregnancy test (urine), and sedimentation rate | Local laboratory | 9.7.5, 9.7.4.1 | | |
| | Phe, phenylalanine; PK, pharmacoki | netic. | | | |
| | <sup>a</sup> Analysis of the anti-rAvPAL-PEG I<br>Organization. | gE assay will be performed by | a Contract Research | | |
| Section 9.7.1.1/<br>Demographic Data and<br>Medical History | Demographic data and a detailed be obtained at Screening. | l medical history <u>, includin</u> | g allergy history, will | | 22 |
| Section 9.7.1.2/<br>Physical Examination | Physical examination will include dermatologic; head, eyes, ears, n | | = = | | 27 |
| Findings | musculoskeletal; and neurologic | | • • • | | |



| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | Screening only. | | |
| Section 9.7.1.3/Vital Sign<br>Measurements | Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, weight (kg), and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. | | 27 |
| Section 9.7.1.5/Chest<br>X-Ray | A chest X-ray will be performed at the Month 12 and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health. | | 23 |
| Section 9.7.2.1/Blood<br>Phenylalanine<br>Concentrations | In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick as outlined in Table 2.1.1. This may be done by the subject at home. Subjects who have their dose frequency increased will have additional Phe assessments performed as outlined in Table 2.1.2 and 2.1.3. | | 27 |
| Section 9.7.3/ Pharmacokinetic Variables | Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentrations (below 120-600480 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks. | | 10, 18 |
| | on the same day each week for 3 consecutive weeks. Subjects who have increased their dose frequency to twice weekly or daily will | | |



| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | have additional PK assessments performed for 5 weeks after the change in dose regimen (refer to Section 12.3.5 and Tables 2.1.2 and 2.1.3). | | |
| Section 9.7.4.1/<br>Pregnancy Testing | Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 2.1.1 and Table 2.1.2). Female subjects with a positive <u>serum</u> pregnancy test at Screening do not meet eligibility criteria for enrollment. | | 27 |
| Section 9.7.4.2/<br>Antibody Testing | Immunoglobulin G (IgG) and M (IgM) antibodies and neutralizing antibodies (NAb) to rAvPAL PEG will be measured using validated immunogeneticity assays at the timepoints indicated in the Schedule of Events (Table 2.1.1). Anti-PEG antibodies will also be measured. Immunogenicity will be assessed by determining antibody response and neutralizing activity with the following measurements: 1) anti-rAvPAL immunoglobulin G (IgG) antibodies, 2) anti-rAvPAL immunoglobulin M (IgM) antibodies, 3) anti-PEG IgG antibodies, 4) anti-PEG IgM antibodies, 5) anti-rAvPAL-PEG immunoglobulin E (IgE) antibodies, and 6) anti-rAvPAL-PEG Enzyme Activity Neutralizing antibodies (NAb). Validated immunogenicity assays will be used per the time points indicated in the Schedule of Events (Table 2.1.1). BioMarin will perform the analysis except for anti-rAvPAL-PEG IgE antibodies, which will be assessed by a Contract Research Organization. | | 14 |



| Section No./Title | Revision | | Comments | Relates to Change No. |
|---|---|---|---|---|
| Section 9.7.5/Clinical | Table 9.7.5.1: Cl | inical Laboratory Tests has been revised to include tests for the | | 8, 27 |
| Laboratory Assessments | Unscheduled Ski | n Reaction visits. In addition, information has been added to | | |
| | indicate that a lo | cal laboratory will perform sedimentation rate analysis and the | | |
| | other laboratory | tests have been revised for accuracy. | | |
| Section 10.1/Adverse | The Investigator | will determine the severity of each AE and will record it on the | | 16 |
| Events | source document | s and AE CRF, using the categories CTCAE v 3 grades defined | | |
| | below. Events th | at are CTCAE grades 4 and 5 are serious events and require | | |
| | completion of bo | th an SAE form and AE eCRF. | | |
| | Grade | Description | | |
| | 1 | <u>Mild</u> | | |
| | 2 | <u>Moderate</u> | | |
| | 3 | Severe | | |
| | 4 | Life threatening or debilitating | | |
| | <u>5</u> | Death related | | |
| | Mild | No limitation of usual activities | | |
| | Moderate | Some limitation of usual activities | | |
| | Severe | Inability to carry out usual activities | | |

**PAL-003** 


| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Section 10.4/BioMarin<br>Pharmacovigilance<br>Contact Information | Contact information for the Mmedical Mmonitor is as follows: Name: Address: Novato, CA 94949 USA Phone: Fax: E-mail: | | 25 |
| Section 12.2/Screening<br>Visit | <ul> <li>Medical history, including allergy history, and demographics</li> <li>Physical examination and height</li> <li>Vital signs, including height and weight</li> <li>Predose bBlood Phe and plasma tyrosine concentration</li> <li>For subjects who participated in PAL-002, these assessments may be the same used for the Week 16 Final Follow up Visit of PAL-002, if they occur within 28 days from Day 1.</li> </ul> | | 22, 27 |
| Section 12.3.1/Day 1 (Week 1) | <ul> <li>Vital signs, including weight</li> <li>Predose PK sample</li> <li>Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)</li> </ul> | | 27 |
| Section 12.3.2/Weekly | Vital signs, including weight | | 15, 20, 27 |


**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| Visits | <ul> <li>3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)</li> <li>Predose PK sample <ul> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 µmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.</li> </ul> </li> <li>Predose blood Phe and plasma tyrosine concentration <ul> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 µmol/L for the majority of the 3 months), the predose plasma Phe and tyrosine assessments may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. The weekly plasma Phe assessment may be replaced with a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes.</li> </ul> </li> </ul> | | |
| Section 12.3.3/Monthly Visits | Monthly visits consist of all weekly activities and include additional activities. The following study activities will be performed at the monthly visits beginning with Week 4: • Vital signs, including weight | | 15, 20, 27 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | <ul> <li>Chest x-ray (Month 12 visit only)</li> <li>3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)</li> <li>Predose PK sample (subjects who are on a stable dosing regimen for ≥3 months only)</li> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 µmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.</li> </ul> | | |
| | <ul> <li>Predose blood Phe and plasma tyrosine concentration</li> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 µmol/L for the majority of the 3 months), the predose plasma Phe and tyrosine assessments may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. The weekly plasma Phe assessment may be replaced with a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes.</li> <li>Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG)</li> </ul> | | |
| | IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE) | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home. | | |
| Section 12.3.4/Quarterly Visits (Week 12, 24, 36, etc.) | <ul> <li>Quarterly visits consist of all weekly and monthly activities and include additional activities. The following study activities will be performed at the quarterly visits beginning with Week 12: <ul> <li>Vital signs, including weight</li> <li>3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)</li> <li>Predose PK sample (subjects who are on a stable dosing regimen for ≥3 months only)</li> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.</li> <li>Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgE)</li> <li>In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.</li> </ul> </li> </ul> | | 15, 20, 27 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| Section 12.3.5/Interim | Subjects who increase their dose frequency from 1x/week to 2x/week or daily will | | 10 |
| Dosing Visit | have additional assessments performed for 5 weeks after the subject's | | |
| | rAvPAL-PEG dose frequency has been increased. If the Interim Dosing Visit | | |
| | coincides with a weekly, monthly, or quarterly scheduled visit, the scheduled visit | | |
| | assessments should also be performed. The following study activities will be | | |
| | performed for the Interim Dosing Visit: | | |
| | • Vital signs, including weight | | |
| | • <u>Injection-site inspection (previous and current injection site)</u> | | |
| | • Assessment of AEs | | |
| | • Concomitant medications | | |
| | Blood Phe measurement by fingerstick | | |
| | o This may be done by the subject at home. | | |
| | • <u>PK sample</u> | | |
| | Subjects who increase their dose frequency to 2x/week will have an additional predose PK sample obtained prior to administration of the first 4 doses (ie, for 2 weeks after the dose frequency increase). For the remaining 3 weeks after the dose frequency increase, a PK sample will be obtained weekly prior to the first dose. Refer to Table 2.1.2 for the Interim Dosing Visit schedule. | | |
| | <ul> <li>Subjects who have their dose frequency increased to daily will have additional PK samples obtained every day for the first week:</li> <li>12 hours after the first daily dose and predose every day for the</li> </ul> | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | rest of the week. After the first week of daily dosing, subjects will have weekly PK samples obtained for 4 additional weeks. Refer to Table 2.1.3 for the Interim Dosing Visit schedule. | | |
| Section 12.3.6/<br>Unscheduled<br>Hypersensitivity Reaction<br>Visit | Subjects who have a generalized skin reaction after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 48 hours) the reaction. Subjects who have other systemic symptoms or a large local skin reaction that is not contiguous to the injection site (refer to Section 9.1.1) may have these assessments performed per investigator discretion. • Injection-site inspection • Clinical laboratory tests • Sedimentation rate • CRP, CH50, C <sub>1</sub> , and C <sub>4</sub> • Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE) • Serum tryptase level • Perform immediately after reaction if possible. • Assessment is optional for subjects who have a generalized skin reaction per investigator discretion. • PK sample | | 8 |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to<br>Change No. |
|---|---|---|---|
| | Assessment of AEs | | |
| | Concomitant medications | | |
| | Subjects should then return to the clinic 4 weeks after their last dose of | | |
| | rAvPAL-PEG for the Early Termination Visit assessments (refer to Section 12.4). | | |
| Section 12.4/Early | 12.4 Final Follow up Visit (Day 113 [±3 days])/Early Termination Visit | | 21, 27 |
| Termination Visit | The final follow up (F/U) Visit or Early Termination Visit (ETV) will occur | | |
| | 4 weeks after the final dose of study drug. | | |
| | Subjects who complete an Unscheduled Hypersensitivity Reaction Visit (refer to | | |
| | Sections 12.3.6) will be terminated from the study. Subjects will then return | | |
| | 4 weeks after the last dose of study drug for the Early Termination Visit. | | |
| | The following study activities will be performed at the F/U Visit or ETV: | | |
| | Physical examination and weight | | |
| | Vital signs, including weight | | |
| | • <u>Chest x-ray</u> | | |
| | • PK sample | | |
| | • Predose bBlood Phe and plasma tyrosine concentration | | |
| | • Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti- | | |

**PAL-003** 

| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | rAvPAL-PEG IgE) | | |
| Section 12.5/Final<br>Follow-up Visit (Day 113<br>[±3 days]) | 12.54 Final Follow-up Visit (Day 113 [±3 days]) /Early Termination Visit Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the | | 21, 27 |
| | ETV will be followed by the Investigator. | | |
| | Every reasonable effort should be made to contact any subject who is lost to follow up. | | |
| | The following study activities will be performed at the F/U Visit or ETV: | | |
| | • Vital signs, including weight | | |
| | • <u>Chest x-ray</u> | | |
| | • PK sample | | |
| | • Predose bBlood Phe and plasma tyrosine concentration | | |
| | Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE) | | |
| Section 14.2/Safety | All subjects who receive any amount of study drug in this study and have | | 19, 27 |
| Analysis | postdose safety information will be included in the safety analyses. | | |
| | Safety will be evaluated on the incidence of AEs, including serious AEs (SAEs), and clinically significant changes in vital signs and laboratory test results. | | |

**PAL-003** 


| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| | The verbatim terms reported on CRFs to identify AEs will be coded using MedDRA. Treatment-emergent AEs will be summarized for each treatment group by system organ class, preferred term, relationship to study drug, and severity. Changes from baseline in vital signs and laboratory test results will be summarized with descriptive statistics by dose group. | | |
| Section 14.3/<br>Pharmacokinetic<br>Analysis | Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (below 120-600480 µmol/L) for a minimum of 2 weeks and no further dose modification is planned. Should data become available from PAL 001 and/or PAL-002 which that indicate study drug accumulation should also be measured, the protocol will be amended to require additional blood draws may be added for PK analysis as needed but not to exceed 3x/week. | | 18, 27 |
| Section 14.4/Efficacy<br>Analysis | In addition, the proportion of subjects who have maintained target Phe concentrations of 120-600 μmol/L will be summarized by each scheduled time point. | | 19 |
| Section 14.7/Interim<br>Analysis | At least one interim analysis may be performed by the sponsor during the study. Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC). | | 27 |
| Section 15/Data<br>Monitoring Committee | The DMC will act <u>independently</u> in an advisory capacity to BioMarin to monitor | | 27 |




| Section No./Title | Revision | Comments | Relates to Change No. |
|---|---|---|---|
| (DMC) | the subjects afety and the efficacy of rAvPAL-PEG in subjects who participate in the study. | | |
| Section 21/References | Burgard, Bremer, Bührdel, Clemens, Mönch, Przyrembel, Trefz, Ullrich. Rationale for the German recommendations for phenylalanine level control in phenylketonuria 1997. Eur J Pediatr 158, 46–54. 1999. Butterworth. Effects of hyperammonaemia on brain function. J Inherit Metab Dis 21 Suppl 1, 6–20. 1998. | | 27 |



## CLINICAL STUDY PROTOCOL

Study Title: Long-term Extension of a Phase 2, Open-Label Dose-

Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of

rAvPAL-PEG in Subjects with PKU

**Protocol Number:** PAL-003

Investigational Product: rAvPAL-PEG
IND/EUDRACT Number: IND 076269

**Indication:** Phenylketonuria

**Sponsor:** BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

**Development Phase:** Phase 2

Sponsor's Responsible

Medical Officer: , Clinical Sciences

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

**Duration: 24 months** or until study is terminated

, MD

**Dose:** 0.001 to 1.0 mg/kg per individual injection, with a

maximum weekly dose of 2.0 mg/kg

Date of Original Protocol: October 08, 2008

Date of Amendment 1: February 09, 2009

Date of Amendment 2: October 30, 2009


 ${\bf May\ not\ be\ divulged,\ published,\ or\ otherwise\ disclosed\ to\ others\ without\ prior\ written}$ 

approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.



#### 2 SYNOPSIS

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


**STUDY SITES:** Approximately 8 centers in the United States

PHASE OF DEVELOPMENT: Phase 2

#### STUDY RATIONALE:

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding study (Study PAL-002). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

#### **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of **multiple doses of** SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.
- To evaluate steady-state PK of rAvPAL-PEG in subjects with PKU.

| BIOMARIN° PAL-003 |
|-------------------|
|-------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### STUDY DESIGN AND PLAN:

This is a long-term extension of a Phase 2, open-label, dose-finding study (Study PAL-002) in 35-50 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002.

Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety as determined by blood Phe concentrations. If a subject's blood Phe concentration is <120  $\mu$ mol/L, the subject's diet may be adjusted to increase the amount of dietary Phe intake to maintain target blood Phe concentrations of 120-600  $\mu$ mol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

At least one interim analysis may be performed by the sponsor during the study. In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 **subjects**' rAvPAL-PEG dosing will continue in PAL-003 without interruption of dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations **of 120-600** μmol/L. **Doses** will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (120-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed but not to exceed 3x/week (fingerstick tests may be performed more frequently).

A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The subject has completed the study through the Month 24 visit.
- 4. The study is terminated.

| BIOMARIN | PAL-003 |
|----------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

### **Dose Modifications:**

After any modifications (increases or decreases) to dose level or frequency, subjects should remain in the clinic for observation for at least 2 hours following the injection of study drug. The Investigator should remain at the site to assess the subject for safety.

#### Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. **Decisions regarding dose increases will depend on blood Phe and drug concentrations**.

Blood Phe levels will be measured 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed.

Depending upon the response to rAvPAL-PEG in PAL-002, **an individual** subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.3, 0.6, and 1.0 mg/kg) that were defined in the previous study (PAL-002).
- The dose\_may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 2.0 mg/kg, including subjects who receive more than 1 dose/week. Subjects who increase their dose frequency will have additional assessments performed (Interim Dosing Visit).
- When a dose is **increased** (either by **increasing** the dose level or by **increasing** the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time.
- Only 1 dose adjustment is allowed every 2 weeks.
- Blood Phe levels will be measured 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed.

## **Dose Decrease Methodology**

A subject's diet should be assessed prior to any dose decreases. Changes to diet should only be made if a subject's blood Phe concentrations <120 μmol/L. If a subject's blood Phe level is

| BIOMARIN PAL-003 |
|-------------------------------|
|-------------------------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

 $<\!120~\mu mol/L$ , the subject's dietary Phe intake should be increased to achieve a stable blood Phe concentration of 120-600  $\mu mol/L$ . If the subject's blood Phe level is  $<\!120~\mu mol/L$  despite a high Phe diet, the rAvPAL-PEG dose will then be decreased. The subject will be asked about any changes to diet prior to any dose adjustments, and any changes to diet should be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (>30% change from baseline) and drug concentrations, as well as toxicity (any hypersensitivity reaction). Dose decreases may occur for safety (ie, blood Phe concentration <120 µmol/L) or other toxicity that may be improved with a lower, more frequent dose.

A dose should first be reduced by dose level (1.0, 0.6, 0.3, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced.

#### Stopping Criteria:

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level.

In addition, if 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater, further dosing of subjects at that dose level will be halted and no subjects will be treated at a higher dose level until a safety assessment is completed. In addition, the Food and Drug Administration (FDA) will be notified of this occurrence.

### **NUMBER OF SUBJECTS PLANNED:**

35-**50** subjects.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in PAL-002.
- 2. Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, during study participation.



| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL-002.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

### INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

rAvPAL-PEG doses will be administered SC and the dosage that provides control of blood Phe concentrations within the target range of 120-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses.

### **DURATION OF TREATMENT:**

Extension of multiple dosing will continue until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The subject has completed the study through the Month 24 visit.
- 4. The study is terminated.



| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

## REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

#### **CRITERIA FOR EVALUATION:**

## **Efficacy:**

Blood Phe concentrations will be measured.

## **Immunogenicity:**

The presence of antibodies will be assessed.

## **Safety:**

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs or laboratory test results.

#### **Pharmacokinetic:**

Plasma concentrations of rAvPAL-PEG will be measured when steady-state levels of Phe are attained.

### STATISTICAL METHODS:

## Sample Size:

Subjects who participated in PAL-002 may be enrolled into this study. No formal sample size calculation was conducted.

#### **Safety Analysis:**

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

Safety will be evaluated on the incidence of AEs, including serious AEs (SAEs), and clinically significant changes in vital signs and laboratory test results.

### **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe

| BIOMARIN | PAL-003 |
|----------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

concentrations of 120-600 µmol/L will be summarized by each scheduled time point.

## Pharmacokinetic Analysis:

Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis.

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (120-600  $\mu$ mol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Should data become available from PAL-002 that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed but not to exceed 3x/week.




## 2.1 Schedule of Events

**Table 2.1.1: Schedule of Events** 

| | | Treatment Period <sup>b,c</sup> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly | Monthly (eg,<br>Wk 4, 8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Final F/U Visit | Early Term.<br>Visit | Unsched.<br>Hyper. |
| Assessments and Events | Screeninga | D 1 | Starting at<br>Week 2 | Every 4th week; Perform in addition to weekly procedures | Every 12th week. Perform in addition to monthly procedures | 1 week after<br>final dose | 4 weeks after final dose | Reaction Visit. <sup>d</sup> Perform within 48 hours; then perform Early Term. procedures |
| Informed consent | X | | | | | | | |
| Medical history, including allergy history, and demographics | X | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | | X | X | X | |
| Vital signs and weight | X | X | X | | | X | X | |
| 12-lead ECG | X | | | | | X | X | |
| Clinical laboratory tests | X | | | X | | X | X | $\mathbf{X}^{\mathbf{g}}$ |
| Sedimentation rate | | X | | | X | X | X | X |
| Chest x-ray | | | | X<br>(12-month<br>visit only) | | X | X | |
| Urine pregnancy test <sup>h</sup> | X | X | | X | | X | X | |
| Injection-site inspection | | X<br>(postdose) | X | | | X | X | X |
| Adverse events <sup>j</sup> | Χ← | | | | | >X | X | X |
| Concomitant medications | X | X | X | | | X | X | X |
| Diet query | X | X | X | | | X | X | |
| 3-Day diet diary <sup>R</sup> | | | X | | | | | |
| Serum rAvPAL-PEG antibodies 1 | | X | | X | | X | X | X |
| Predose <b>plasma</b> Phe and plasma tyrosine <sup>m</sup> | X | X | X <sup>n</sup> | | | X<br>(postdose) | X<br>(postdose) | |
| Plasma Phe (fingerstick) <sup>6</sup> | | | (3 days<br>postdose) | | | | | |
| Plasma PK sample <sup>p</sup> | | X | X <sup>n</sup> | | | X | X | X |
| Administer IP <sup>q</sup> | | X | X | | | | | |
| Serum tryptase level <sup>r</sup> | | | | | | | | X |

| BIO | M | A | R | N | 9 |
|-----|---|---|---|---|---|
|-----|---|---|---|---|---|


AE, adverse event; **CH50, total hemolytic complement; CRP, C-reactive protein;** D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; **Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M;** IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

- <sup>a</sup> It is preferable to perform PAL-003 Screening assessments the same day as PAL-002 **Week 16 visit** so there is no interruption of study drug. If performed on the same day, PAL-002 **Week 16 visit** data may be used. If not, PAL-003 Day 1 must occur ≤ 28 days after PAL-003 Screening.
- <sup>b</sup> Additional visits may occur if deemed necessary to monitor AEs or blood Phe, adjust dosing etc.
- <sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.
- <sup>d</sup> Unscheduled hypersensitivity reaction assessments are mandatory for subjects who have a generalized skin reaction. Subjects who have other systemic symptoms or who have a large local skin reaction that is not contiguous to the injection site may have these assessments performed per investigator discretion. Assessments should be performed within 48 hours of the reaction. Subjects who complete an Unscheduled Hypersensitivity Reaction Visit must be terminated from the study and should complete an Early Termination Visit.
- <sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.
- <sup>f</sup> Clinical laboratory tests to include hematology, chemistry, and urinalysis.
- g Subjects who have a generalized skin reaction should also be assessed for CRP, CH50, C<sub>1</sub>, and C<sub>4</sub> within 48 hours of the reaction. Subjects who have other systemic symptoms or who have a large local skin reaction that is not contiguous to the injection site may have these assessments performed per investigator discretion.
- <sup>h</sup> If positive or equivocal, perform serum pregnancy test.
- <sup>i</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, e.g. right arm vs. left arm).
- <sup>j</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug to the final study visit.
- <sup>k</sup> It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.
- <sup>1</sup> Includes testing for anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE antibodies.
- <sup>m</sup> Samples should be drawn in the morning, at least 2.5 hours after a meal. **If dose is modified by increasing dose level, additional blood Phe concentration testing should be done on the third day following dose adjustment.** If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.
- <sup>n</sup> Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose plasma Phe, tyrosine, and PK assessments may be skipped at the weekly visits and performed at the monthly visits for




the first year then 2-3 months thereafter. The weekly plasma Phe assessment may be replaced by a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes.

- <sup>o</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.
- <sup>p</sup> The PK blood samples will be collected after the subject has achieved and maintained target blood Phe concentrations (120-600 μmol/L) for a minimum of 2 weeks. Once this target is achieved, predose PK samples will be collected on the same day each week for 3 consecutive weeks.
- <sup>q</sup> Dosing is up to 1.0 mg/kg per injection and up to one dose per day, for a total **not to exceed** 2.0 mg/kg/week, **including subjects who receive more than 1 dose/week**. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency will need to be re-evaluated.
- <sup>r</sup> Mandatory for subjects who have a large local skin reaction that is not contiguous to the injection site or non-skin systemic symptoms. Optional for subjects who have a generalized skin reaction. Take sample immediately after reaction if possible.




Table 2.1.2: Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to 2x/Week

| | | | S | ubjects Who | Are Administe<br>Treatmen | | -PEG 2x/Wee | k | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | First Week After Dose Adjustment Second Week After Dose Adjustment Adjustment Adjustment | | | | | | _ 0 0== 0== | eek After<br>justment | Fifth Week After Dose<br>Adjustment | |
| Assessments and Events | First Dose | Second<br>Dose | First Dose | Second<br>Dose | First Dose | Second<br>Dose | First Dose | Second<br>Dose | First Dose | Second<br>Dose |
| Vital signs and weight | X | X | X | X | X | X | X | X | X | X |
| Injection-site inspection | X | X | X | X | X | X | X | X | X | X |
| Adverse events <sup>c</sup> | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X |
| Plasma PK sample | X | X | X | X | X | | X | | X | |
| Blood Phe (fingerstick) <sup>d</sup> | X | X | X | X | X | X | X | X | X | X |

AE, adverse event; D, day; PK, pharmacokinetics; Phe, phenylalanine.

<sup>&</sup>lt;sup>a</sup> The additional Interim Dosing Visit assessments should be performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased to 2x/week. All assessments should be performed predose unless specified otherwise.

<sup>&</sup>lt;sup>b</sup> If the Interim Dosing Visit coincides with a regularly scheduled visit, the scheduled visit assessments should also be performed.

<sup>&</sup>lt;sup>c</sup> If any injection site reaction is observed, the corresponding AE data must specify injection location (identify current vs. previous visit's injection, e.g., right arm vs. left arm).

<sup>&</sup>lt;sup>d</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.




Table 2.1.3: Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to Daily

| | | Sub | jects Who Are Adminis<br>Treatment | | aily | |
|---|---|---|---|---|---|---|
| | First Day After<br>Dose Adjustment | First Week After<br>Dose Adjustment | Second Week After<br>Dose Adjustment | Third Week After<br>Dose Adjustment | Fourth Week After<br>Dose Adjustment | Fifth Week After<br>Dose Adjustment |
| Assessments and Events | Dose 1 | Doses 2-7 | Doses 8-14 | Doses 15-21 | Doses 22-29 | <b>Doses 30-36</b> |
| Vital signs and weight | X | X | X | X | X | X |
| Injection-site inspection | X | X | X | X | X | X |
| Adverse events <sup>c</sup> | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X |
| Plasma PK sample | X<br>(12 hours postdose) | X<br>(Daily) | 1x/week | 1x/week | 1x/week | 1x/week |
| Blood Phe (fingerstick) <sup>d</sup> | X | X | X | X | X | X |

AE, adverse event; D, day; PK, pharmacokinetics; Phe, phenylalanine.

<sup>&</sup>lt;sup>a</sup> The additional Interim Dosing Visit assessments should be performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased to daily. All assessments should be performed predose unless specified otherwise.

<sup>&</sup>lt;sup>b</sup> the Interim Dosing Visit coincides with a regularly scheduled visit, the scheduled visit assessments should also be performed.

<sup>&</sup>lt;sup>c</sup> If any injection site reaction is observed, the corresponding AE data must specify injection location (identify current vs. previous visit's injection, e.g., right arm vs. left arm).

<sup>&</sup>lt;sup>d</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.




# **3 TABLE OF CONTENTS**

| 1 | TITLE PAGE | 1 |
|---|-------------------------------------------------------------------|-----|
| 2 | SYNOPSIS | 2 |
| | 2.1 Schedule of Events | |
| 3 | TABLE OF CONTENTS | 15 |
| 4 | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 19 |
| 5 | ETHICS | 23 |
| | 5.1 Institutional Review Board or Ethics Committee | 23 |
| | 5.2 Ethical Conduct of Study | 23 |
| | 5.3 Subject Information and Informed Consent | |
| 6 | INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE | 25 |
| 7 | INTRODUCTION | 26 |
| | 7.1 Nonclinical Studies | 26 |
| | 7.2 Previous Clinical Studies | 28 |
| | 7.3 Study Rationale | 28 |
| | 7.4 Summary of Overall Risks and Benefits | 29 |
| | 7.4.1 Toxicity Due to Exposure to PEG | 29 |
| | 7.4.2 Toxicity Due to an Immunologic Reaction | 30 |
| | 7.4.3 Effects of Low Blood Phe | 33 |
| 8 | STUDY OBJECTIVES | 34 |
| 9 | INVESTIGATIONAL PLAN | 35 |
| | 9.1 Overall Study Design and Plan | 35 |
| | 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEC | i36 |
| | 9.1.2 Dose Modifications | 41 |
| | 9.1.3 Stopping Criteria | 42 |
| | 9.2 Discussion of Study Design, Including Choice of Control Group | 43 |
| | 9.3 Selection of Study Population | |
| | 9.3.1 Inclusion Criteria | 43 |
| | 9.3.2 Exclusion Criteria | 43 |




| | 9.3.3 | Removal of Subjects from Treatment or Assessment | 44 |
|----|------------|----------------------------------------------------|----|
| | 9.3.4 | Subject Identification and Replacement of Subjects | 45 |
| | 9.4 Trea | itments | |
| | 9.4.1 | Treatments Administered | 46 |
| | 9.4.2 | Identity of Investigational Product (IP) | 46 |
| | 9.4.3 | Storage | 46 |
| | 9.4.4 | Directions for Administration | 46 |
| | 9.4.5 | Method of Assigning Subjects to Treatment Groups | 48 |
| | 9.4.6 | Selection of Doses Used in the Study | 48 |
| | 9.4.7 | Blinding | 49 |
| | 9.4.8 | Prior and Concomitant Medications | 49 |
| | 9.4.9 | Treatment Compliance | 50 |
| | 9.5 Inve | estigational Product Accountability | 50 |
| | 9.5.1 | Return and Disposition of Clinical Supplies | 50 |
| | 9.6 Diet | ary or Other Protocol Restrictions | 50 |
| | 9.7 Effic | cacy and Safety Variables | 51 |
| | 9.7.1 | Efficacy and Safety Measurements Assessed | 51 |
| | 9.7.2 | Efficacy Variable | 52 |
| | 9.7.3 | Pharmacokinetic Variables | 52 |
| | 9.7.4 | Safety Variables | 53 |
| | 9.7.5 | Clinical Laboratory Assessments | 53 |
| 10 | REPORT | ING ADVERSE EVENTS | 56 |
| | 10.1 Adv | erse Events | 56 |
| | 10.2 Serie | ous Adverse Events | 59 |
| | 10.3 Preg | nancy | 60 |
| | 10.4 Biol | Marin Pharmacovigilance Contact Information | 60 |
| 11 | APPROPI | RIATENESS OF MEASUREMENTS | 61 |
| | 11.1 Safe | ety and Pharmacokinetics | 61 |
| 12 | | PROCEDURES | |
| | 12.1 Pres | tudy | 61 |

| BIOI | MA | RI | N |
|------|----|----|---|
|------|----|----|---|


| | 12.2 Screening Visit | 61 |
|----|--------------------------------------------------------------|----|
| | 12.3 Treatment Period | 62 |
| | 12.3.1 Day 1 (Week 1) | 62 |
| | 12.3.2 Weekly Visits | 63 |
| | 12.3.3 Monthly Visits (Week 4, 8, 12, etc) | 63 |
| | 12.3.4 Quarterly Visits (Week 12, 24, 36, etc) | 65 |
| | 12.3.5 Interim Dosing Visit | 66 |
| | 12.3.6 Unscheduled Hypersensitivity Reaction Visit | 66 |
| | 12.4 Early Termination Visit | 68 |
| | 12.5 Final Follow-up Visit | 69 |
| 13 | DATA QUALITY ASSURANCE | 70 |
| 14 | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 71 |
| | 14.1 Statistical and Analytical Plans | 71 |
| | 14.2 Safety Analysis | 71 |
| | 14.3 Pharmacokinetic Analysis. | 71 |
| | 14.4 Efficacy Analysis | 71 |
| | 14.5 Determination of Sample Size | 72 |
| | 14.6 Handling of Missing Data | 72 |
| | 14.7 Interim Analyses | 72 |
| | 14.8 Changes in the Conduct of the Study or Planned Analyses | 72 |
| 15 | DATA MONITORING COMMITTEE (DMC) | 74 |
| 16 | COMPENSATION, INSURANCE, AND INDEMNITY | 75 |
| 17 | CASE REPORT FORMS AND SOURCE DOCUMENTS | 76 |
| 18 | STUDY MONITORING AND AUDITING | 78 |
| 19 | RETENTION OF RECORDS. | 79 |
| 20 | USE OF INFORMATION AND PUBLICATION | 80 |
| 21 | REFERENCES | 81 |
| 22 | INVESTIGATOR RESPONSIBILITIES | 83 |
| | 22.1 Conduct of Study and Protection of Human Subjects | 83 |




# LIST OF TABLES

| Table 2.1.1: Schedule of Events | 10 |
|---|---|
| Table 2.1.2: Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to 2x/Week | 13 |
| Table 2.1.3: Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to Daily | 14 |
| Table 9.4.4.1 Number of Injections Required For an Individual Weighing 80 kg | 48 |
| Table 9.7.1.1: Summary of Laboratory Assessments | 51 |
| Table 9.7.5.1: Clinical Laboratory Tests | 55 |

## LIST OF FIGURES




### 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

## **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

AUC<sub>0-7 days</sub> area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen

°C degree Celsius

**CBC** complete blood count

CD Compact disk

CFR Code of Federal Regulations
CH50 total hemolytic complement

C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form
CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure
DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up

g gram

GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal




IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IgEimmunoglobulin EIgGimmunoglobulin GIgMimmunoglobulin MIPinvestigational productIRBInstitutional Review Board

IV intravenous kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hgmillimeter of mercuryNAbneutralizing antibodiesNCINational Cancer Institute

NOAEL no observable adverse effect level

OTC over the counter

PAH phenylalanine hydroxylase PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator
PK pharmacokinetics
PKU phenylketonuria

rAvPAL-PEG rAv phenylalanine ammonia lyase-PEG

RBC red blood cell

SAE serious adverse event
SAP Statistical Analysis Plan
SBP systolic blood pressure

SC subcutaneous

SD standard deviation



SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase SGPT serum glutamic pyruvate transaminase

US United States
WBC white blood cell


## Definition of Terms:

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.



### 5 ETHICS

## 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

# 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will



provide written, informed consent before any study-related tests or evaluations are performed.

## 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR §50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



## 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Regulatory Affairs Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.



### 7 INTRODUCTION

A comprehensive review of phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

## 7.1 Nonclinical Studies

The murine model of phenylketonuria (PKU) BTBRPah<sup>enu2</sup> (ENU2), a mouse line that is deficient in phenylalanine hydroxylase (PAH) activity (Shedlovsky, 1993, Genetics), was used for in vivo screening and pharmacodynamic studies. This mouse model exhibits characteristics similar to those seen in PKU patients, including hyperphenylalaninemia (baseline plasma phenylalanine [Phe] concentrations of 1000 to 2000 µM) and hypopigmentation. Weekly subcutaneous (SC) administration of 80 mg/kg of rAvPAL-PEG (approximately 4 IU/mouse) for greater than 2 to 3 months lowered and stabilized plasma Phe concentration from approximately 2000 µM to less than 200 µM. A similar profile of Phe reduction was also seen in ENU2 mice administered wild-type AvPAL-PEG (4 IU/mouse) over 8 weeks. In all these studies, regardless of the molecule, an attenuated Phe-lowering response was usually seen between Weeks 2 and 7. However, plasma Phe concentrations became stable at concentrations below 200 µM from Week 7 onward. In addition to the reduction of plasma Phe, a dose-related darkening in coat color occurred, indicating the biosynthesis of melanin, which was previously inhibited when plasma Phe could not be metabolized and plasma Phe concentrations were high. When administration of AvPAL-PEG was stopped for 2 to 7 weeks and then reinitiated with weekly administrations, no attenuated response was observed and Phe concentrations remained low and stable until the next administration.

The safety of rAvPAL-PEG was evaluated in safety pharmacology studies (respiratory, central nervous system [CNS] and cardiovascular [CV]) and toxicity with toxicokinetic studies (single and 28-day repeated dose) in rats and cynomolgus monkeys. Overall, in **the nonclinical** studies, no **anaphylactoid-like reactions or injection-site reactions were noted.** No specific polyethylene glycol (PEG)-related histological findings were observed during the 28-day repeated dose studies.

Findings in cynomolgus monkeys dosed with a single administration of 60 mg/kg rAvPAL-PEG included reduced food consumption, dehydration, body weight loss, hypoactivity, hypothermia, decreased plasma Phe concentration, decreased protein synthesis, and gastrointestinal (GI) lesions. Plasma Phe concentrations were also reduced to below the



**PAL-003** 


level of detection in the 4 and 12 mg/kg dose groups, but without similar toxicological consequences, implying that the physiological regulation of Phe levels may be an important factor for influencing morbidity.

The main finding in the 28-day study was the possible drug-related observation of minimal to slight degeneration of blood vessels of predominantly medium-sized muscular arteries with a non-dose-dependent involvement of different organs observed in 1 male in the 0.1 mg/kg and 1 male and 1 female in the 1.0 mg/kg rAvPAL-PEG dose groups. No degeneration of the arteries was observed in **either the control or** animals administered 0.01 mg/kg rAvPAL-PEG.

The half-life of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg, was 47, 33, and 44 hours, respectively, and exhibited modest area under the plasma concentration-time curve (AUC)-dose linearity. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the half-life was 65 hours at 4 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum plasma concentration, along with a long half-life, (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) AUC and the maximum plasma concentration (C<sub>max</sub>) are roughly linearly proportional.

Chronic repeat-dose toxicity and toxicokinetic studies were conducted in the rat (17/26 weeks) and monkey (39 weeks). In the 26-week study of rats, weight loss was observed in the rats given 25 mg/kg/dose of rAvPAL-PEG, SC; corresponding decreased food consumption was observed in the males. The main histological finding was focal-to-multifocal areas of vacuolar degeneration of renal tubule cells in the kidney of 3 males given 25 mg/kg and 3 females given  $\geq 8$  mg/kg rAvPAL-PEG. This renal tubule finding persisted in the kidney of both sexes given  $\geq 8$  mg/kg/dose at the end of the 12-week recovery phase without evidence of reversibility. Increased vacuolation was observed in histiocytic cells of the liver, spleen, mesenteric lymph node, mandibular lymph node, and adrenal cortex of males given 25 mg/kg/dose and females given  $\geq 8$  mg/kg/dose; vacuolation of histiocytic cells in the testes were also observed in males given 25 mg/kg/dose. Both renal tubule vacuolation and histiocytic cell vacuoles

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

have been associated with PEG-related catabolism and administration of other PEGylated proteins.

In the 39-week, chronic repeat-dose toxicity and toxicokinetic study in monkeys, dose levels of 7.0 and 5.0 mg/kg/dose rAvPAL-PEG were not tolerated in female monkeys and resulted in body weight loss, decreased food consumption, and hypoactivity. The only adverse microscopic finding was arterial inflammation of small and mid-sized arteries in multiple organs and/or tissues in most animals that were given ≥3 mg/kg/dose rAvPAL-PEG SC twice weekly at the end of the dosing phase. The inter-individual organ involvement was highly variable; some animals had findings in one organ and others had multiple organs with arterial inflammation. Additionally, not all arteries had signs of inflammation and arterial inflammation was resolved by the end of the 13-week recovery period. A full analysis of these findings including the involvement of the anti-drug antibodies, antibody isotypes, PEG distribution, and rAvPAL-PEG is ongoing. The no observable adverse effect level (NOAEL) for the 17-week and 39-week studies, in rat and monkey, respectively, is 1 mg/kg/dose. The NOAEL from these studies represents greater than a 100-fold safety factor over the starting dose in PAL-002.

## 7.2 Previous Clinical Studies

This study is an extension of the second human clinical study with rAvPAL-PEG (Study PAL-002). Study PAL-001, the first-in-human clinical study of rAvPAL-PEG, was designed as a Phase 1, open-label, single-dose, dose-escalation study in 25 subjects, 16 to 50 years old, with PKU. The doses for this study are based on data from nonclinical studies and PAL-001 and are 0.001 through 1.0 mg/kg per injection (not to exceed 2.0 mg/kg/week, provided no dose-limiting toxicity was observed in Study PAL-002.

## 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH (Scriver CR, 2001, McGraw-Hill). Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver CR, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver CR, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated 



**PAL-003** 


Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan<sup>®</sup> is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding study (PAL-002). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

# 7.4 Summary of Overall Risks and Benefits

It is not expected that data from PAL-002 will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

## 7.4.1 Toxicity Due to Exposure to PEG

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least



80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given **a single dose of** up to 60 mg/kg rAvPAL-PEG **SC**.

In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

# 7.4.2 Toxicity Due to an Immunologic Reaction

The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylation does not eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing the immunogenicity of the molecule, it is reasonable to expect that some individuals may exhibit immune responses upon exposure to the drug. These immune responses may be clinically irrelevant, cause symptoms of various degrees, or lead to neutralization of biological activity. Subjects participating in clinical trials will be monitored closely with specific antibody titers, sedimentation rates, and complete blood counts (CBCs).

PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.) (Harris, 2003, Nat.Rev.Drug Discov.), however, antibodies against PEG may form when PEG is bound to compounds. (Harris, 2003, Nat.Rev.Drug.Discov.) (Richter, 1983, Int.Arch.Allergy Appl.Immunol.) In some instances, development of such antibodies did not result in any significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.). Administration of rAvPAL-PEG may lead to anti-PEG antibody formation, and the duration of this possible effect is not known. This\_may limit a subject's future ability to be treated with other PEG-containing (eg, Depo-Provera) or PEGylated

(eg, PEG-interferon) injectable drugs. It is therefore recommended that any



PEG-containing injectable drug administered to subjects after completion of this study be done under medical observation.

## 7.4.2.1 Systemic Skin Reactions

Two subjects who were enrolled in Study PAL-001 and received the protocol-defined single dose of rAvPAL-PEG reported systemic skin reactions (generalized skin rash) that were attributed to treatment with study drug. One subject received a single dose of 0.001 mg/kg rAvPAL-PEG, and the other subject received a single dose of 0.01 mg/kg rAvPAL-PEG. Both of these events were reported as serious and followed administration of Depo-Provera injections (medroxyprogesterone injection), an injectable contraception. These allergic reactions are thought to be related to the PEG molecules that are found in both the study drug, rAvPAL-PEG, and Depo-Provera. These reactions are not likely to be experienced concurrent with other birth control medications.

The 2 subjects were administered study drug during PAL-001 and then experienced an allergic reaction following an injection of Depo-Provera. The symptoms of the reactions were hives on the arms and legs and difficulty breathing. The symptoms for both subjects resolved within 1 day following treatment with medication, including the

Depo-Provera was administered participation in PAL-001. A skin prick test with Depo-Provera was administered as part of this examination. One subject had a mild allergic reaction to the test; however, no further reactions or complications were reported following subsequent administration of a full dose of Depo-Provera. The subject continues to receive regular doses (every 3 months) of Depo-Provera, and no further reactions have been reported to date (15OCT2009). The second subject also had a positive reaction to Depo-Provera following administration of the skin prick test. When a subsequent full dose of Depo-Provera was administered, developed hives, itching, and chills. The subject's symptoms resolved within 1 day of taking medication prescribed by an allergist.

The active drug substance in rAvPAL-PEG is a bacterial protein that may elicit immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and others. It is possible that the physio-chemical properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG. Although results from nonclineal studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys did not indicate signs of immune-mediated toxicities, it is possible that the physio-chemical



properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG in humans. It is currently unknown whether administration of PEG-containing drugs, such as Depo-Provera, has a sensitizing effect to PEG in rAvPAL-PEG when administered in humans. Because the exact basis for these reported events and their duration is not known, the use of PEG-containing injectable drugs prior to, during, and after this study is prohibited as a precautionary measure (refer to Sections 9.3.2 and Section 9.4.8.).

# 7.4.2.2 Management of Allergic Reactions

Allergic reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 2 hours post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of allergic reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection.

In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for antibody testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of allergic symptoms:

- Clearing the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. Acetaminophen or ibuprofen (5-10 mg/kg) may also be administered. An allergy and/or immunology consultation should be sought if necessary. Information regarding the management of local skin, large local skin, and systemic



reactions is provided in Section 9.1.1. Detailed instructions for the management of allergic reactions are provided in the Study Reference Manual.

### 7.4.3 Effects of Low Blood Phe

Insufficient Phe intake or excessive rAvPAL-PEG exposure may cause blood Phe concentrations to be too low (eg, < 30  $\mu$ mol/L). Prolonged low blood Phe concentrations can result in a catabolic state associated with poor growth and altered body functions, including mental and physical alterations, loss of appetite, anemia, rashes, and diarrhea. To ensure safety during this study, subjects will be monitored closely with frequent blood Phe concentration determinations. If a subject's blood Phe concentration is too low, the subject's diet, current dose of study drug, or both may be adjusted.



## 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of **multiple doses of** SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.
- To evaluate steady-state PK of rAvPAL-PEG in subjects with PKU.



## 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of a Phase 2, open-label, dose-finding study (PAL-002) in 35-50 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 (0.001 through 1.0 mg/kg per injection), provided no dose-limiting toxicity was observed in PAL-002.

Only subjects who completed participation in PAL-002 will be enrolled into this study. Diet will not be altered during the course of this study, except as necessary for safety as determined by blood Phe concentrations. If a subject's blood Phe concentration is <120 µmol/L, the subject's diet may be adjusted to increase the amount of dietary Phe intake to maintain target blood Phe concentrations of 120-600 µmol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. For information regarding changes to diet for safety and decreases in dose, refer to Section 9.1.2.2.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

At least one interim analysis may be performed by the sponsor during the study. In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 **subjects**' rAvPAL-PEG dosing will continue in PAL-003 without interruption of dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations **of 120-600** µmol/L. **D**oses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 2.1.1, Schedule of Events. After the subject's blood Phe concentration has been controlled to within a target range (120-600 μmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed but not to exceed 3x/week (fingerstick tests may be performed more frequently).



A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The subject has completed the study through the Month 24 visit.
- 4. The study is terminated.

# 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEG

# 9.1.1.1 Subjects Who Have Had Previous Hypersensitivity Reactions to rAvPAL-PEG or a PEG-containing Product

Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from PAL-002 are excluded from participation in this study. Subjects who experienced a generalized skin rash are included in this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in PAL-002 are eligible to participate in this study. Subjects may develop systemic, large local skin, or local skin reactions after enrollment in PAL-003. Refer to Section 9.1.1.2 for definitions of systemic and local skin reactions. For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.

# 9.1.1.2 Definition of Hypersensitivity Reactions to rAvPAL-PEG Administered Subcutaneously

During Study PAL-003, subjects may experience hypersensitivity reactions to rAvPAL-PEG. The hypersensitivity reactions are defined as follows:

Local skin reaction:

• Skin signs or symptoms in 1 affected primary location, ie, hives, wheals, or swelling or an area of erythema, redness, induration, pain, or itching at or near the site of injection.

## Large local skin reaction:

• Skin signs or symptoms, ie, hives, wheals, or swelling or an area of erythema, redness, or induration with pain or itching that extends beyond the site of injection by approximately 6 inches (15 cm) and/or signs or symptoms that are not contiguous to the injection site. These may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure and, therefore, will be managed as a systemic reaction when not contiguous to the injection site.

Systemic reaction (including generalized skin symptoms):



• Skin and non-skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological.

For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.



**B**OMARIN

PAL-003






#### 9.1.1.3.1 Local Skin Reactions

Subjects who have had a local skin reaction (refer to Section 9.1.1.2 for definition) after administration of rAvPAL-PEG in PAL-001, PAL-002, or this study may be premedicated with acetaminophen and antihistamines 1 hour prior to study drug dosing. Recommended premedications are acetaminophen and antihistamine (Zyrtec [cetirizine] is preferred). The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg Zyrtec or 25 to 50 mg oral Benadryl [diphenahydramine]). Because Benadryl can cause drowsiness, it should be administered only if the subject is accompanied by a designated driver.

Symptoms of local reactions may be treated with local application of ice and non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.2.2).

If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

## 9.1.1.3.2 Large Local Skin Reactions

Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be contiguous to the rAvPAL-PEG injection site. The location of the large local skin reaction relative to the rAvPAL-PEG injection site will determine if a subject may remain in the study and continue to be administered rAvPAL-PEG. An example of a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk.

Subjects who have large local skin reactions that are contiguous to the injection site may remain in the study. Subjects who have large local skin reactions that are not contiguous to the injection site may have additional assessments performed (Unscheduled Hypersensitivity Reaction Visit) per Investigator discretion and must then be terminated from the study. A decision to terminate a subject from the study must be agreed to by both the Investigator and the Sponsor's Medical Officer.

## 9.1.1.3.2.1 Large Local Skin Reactions Contiguous to Injection Site

Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may



remain in the study. Large local skin reactions that are contiguous to the injection site should be managed as local skin reactions (refer to Section 9.1.1.3.1). For the remainder of the study, subjects must be premedicated orally with acetaminophen and antihistamines 1 hour prior to study drug dosing. Recommended premedications are acetaminophen and antihistamine (Zyrtec [cetirizine] is preferred). The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg Zyrtec or 25 to 50 mg Benadryl [diphenahydramine]). Because Benadryl can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver.

Symptoms of large local skin reactions may be treated with local application of ice and topical, or all or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

# 9.1.1.3.2.2 Large Local Skin Reactions Not Contiguous to Injection Site

Large local skin reactions that are not contiguous to the injection site may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure to rAvPAL-PEG and, therefore, will be managed as a systemic reaction. Subjects who develop large local skin reactions that are not contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may not continue to participate in the study. Subjects may have additional assessments performed (ie, Unscheduled Hypersensitivity Skin Reaction Visit) immediately after the reaction (within 48 hours): serum anti-rAvPAL-PEG antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL immunoglobulin M [IgM], anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG immunoglobulin E [IgE]); serum tryptase level; sedimentation rate; C-reactive protein (CRP), total hemolytic complement (CH50), and complements C<sub>1</sub> and C<sub>4</sub>; and clinical laboratory tests (urinalysis, chemistry, hematology). Subjects will then be terminated from the study and should be scheduled to complete the Early Termination Visit (refer to Section 12.4).

Symptoms of large local skin reactions may be treated with local application of ice and topical, or al, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

## 9.1.1.3.3 Systemic Reactions

Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a definition) after administration of rAvPAL-PEG will be terminated from the study. Subjects who experience generalized skin symptoms are included in this category. Immediately after the systemic reaction (within 48 hours), subjects with generalized skin symptoms must have additional assessments performed for safety (ie, Unscheduled Hypersensitivity



Skin Reaction Visit): serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE); serum tryptase level (optional; it is recommended that this sample be drawn immediately after reaction); sedimentation rate; CRP, CH50, C<sub>1</sub>, and C<sub>4</sub>; and clinical laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1). Subjects who have a systemic reaction without generalized skin symptoms may have these assessments performed per Investigator discretion. Subjects will then be terminated from the study and should be scheduled to complete the Early Termination Visit (refer to Section 12.4).

## 9.1.2 Dose Modifications

After any modifications (increases or decreases) to dose level or frequency, subjects should remain in the clinic for observation for at least 2 hours following the injection of study drug. The Investigator should remain at the site to assess the subject for safety.

# 9.1.2.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. **Decisions regarding dose increases will depend on blood Phe and drug concentrations**.

Depending upon the response to rAvPAL-PEG in PAL-002, an individual subject's dose may be adjusted beginning on Day 1 of PAL-003 as follows:

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.3, 0.6, and 1.0 mg/kg) that were defined in the previous study (PAL-002).
- The dose\_may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 2.0 mg/kg, including subjects who receive more than 1 dose/week. Subjects who increase their dose frequency should perform the Interim Dosing Visit assessments (refer to Section 12.3.5 and Table 2.1.2 and Table 2.1.3).
- When a dose is **increased** (either by **increasing** the dose level or by **increasing** the frequency of dosing), the subject must remain in the clinic for a minimum of 2 hours following the first modified dose administration, and an Investigator will remain on site during this time.
- Only 1 dose adjustment is allowed every 2 weeks.



• Blood Phe levels will be measured 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed.

## 9.1.2.2 Dose Decrease Methodology

A subject's diet should be assessed prior to any dose decreases. Changes to diet should only be made if blood Phe concentrations are <120  $\mu$ mol/L. If a subject's blood Phe level is <120  $\mu$ mol/L, the subject's dietary Phe intake should be increased to achieve a stable blood Phe concentration of 120-600  $\mu$ mol/L. If the subject's blood Phe level is <120  $\mu$ mol/L despite a high Phe diet, the rAvPAL-PEG dose will then be decreased. The subject will be asked about any changes to diet prior to any dose adjustments, and any changes to diet should be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (>30% change from baseline) and drug concentrations, as well as toxicity (any hypersensitivity reaction as defined in Section 9.1.1.2). Dose decreases may occur for safety (ie, blood Phe concentration <120 µmol/L) or other toxicity that may be improved with a lower, more frequent dose.

A dose should first be reduced by dose level (1.0, 0.6, 0.3, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced.

## 9.1.3 Stopping Criteria

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principle Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study, restart dosing at the same dose level, or restart dosing at a lower dose level.

In addition, if 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater, further dosing of subjects at that dose level will be halted and no subject will be treated at a higher dose level until a safety assessment is completed. In addition, the Food and Drug Administration (FDA) will be notified of this occurrence.



## 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

# 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in PAL-002.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.



- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL-002.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

# 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study at any time without prejudice. The Investigator must withdraw from the study any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:



- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).

If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

# 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in PAL-002. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.



### 9.4 Treatments

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site with a supply of IP sufficient for the completion of the study.

## 9.4.2 Identity of Investigational Product (IP)

# 9.4.2.1 Product Characteristics and Labeling

The rAvPAL-PEG drug product for SC injection is formulated and supplied as a sterile aqueous (colorless to pale yellow) solution in clear, single-use, type-1 borosilicate glass vials. Each 3 mL vial contains  $1.5\pm0.2$  mL to deliver 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with  $1.5\pm0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Dilution instructions are provided in a separate instruction manual.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

Drug product packaging will be identified with the lot number and expiration date, and will be provided in a box labeled with the study number.

## 9.4.3 Storage

At the study site, all IP must be stored at  $5\pm3^{\circ}$ C ( $41\pm5^{\circ}$ F) under the conditions specified in the IB in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 2 mg/kg.

Dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous



measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

The injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). The number of injections required for an individual weighing 80 kg (about 176 pounds) is provided in Table 9.4.4.1 as an example. Note this table is for example purposes only. Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff or other qualified and trained study personnel.



Table 9.4.4.1 Number of Injections Required For an Individual Weighing 80 kg

| Dose Group<br>(mg/kg) | Weight (kg) | Volume of Study Drug (mL) <sup>a</sup> | No. of<br>Injections <sup>b</sup> |
|---|---|---|---|
| 0.001 | 80 | 0.8 | 1 |
| 0.003 | 80 | 0.6 | 1 |
| 0.01 | 80 | 0.8 | 1 |
| 0.03 | 80 | 0.2 | 1 |
| 0.06 | 80 | 0.5 | 1 |
| 0.1 | 80 | 0.8 | 1 |
| 0.3 | 80 | 2.4 | 2 |
| 0.6 | 80 | 4.8 | 2 or 3 |
| 1.0 | 80 | 8.0 | 4 |

<sup>&</sup>lt;sup>a</sup>Study drug is supplied at a concentration of 10 mg/mL and is then diluted by differential amounts as specified in the PAL-003 Pharmacy Manual. Volume to be injected is calculated based on a starting volume attained following dilution.

Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency will need to be re-evaluated.

### 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in PAL-002.

## 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to **120-600** µmol/L will be determined for each subject.

The doses for this study are based upon the results of nonclinical studies and PAL-001. The no observable adverse effect level (NOAELs) from nonclinical studies in rats and

<sup>&</sup>lt;sup>b</sup>Number of injections per dose is dependent upon site policy for SC injections. The number of injections may vary at the discretion of the Investigator.



**PAL-003** 


monkeys represents a greater than 100-fold safety factor over the starting dose administered in PAL-002 (0.001 mg/kg).

## 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered in the morning by clinic staff or other qualified and trained study personnel.

## 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the medical monitor must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in PAL-002) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior **local skin** reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and antihistamines (refer to Section 9.1.1). If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior **systemic** reaction to rAvPAL-PEG or a PEG-containing product **are excluded from participation in this study** (refer to Section 9.1.1).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.



## 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

# 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

# 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

### 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study except as necessary for safety. If a subject's blood Phe concentration is <120 µmol/L, the subject's diet will be adjusted to maintain blood Phe concentrations of 120-600 µmol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record



immediately prior to their next dose of study drug. The dietary record will be maintained with the study source documents.

## 9.7 Efficacy and Safety Variables

## 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis (Section 2.1) describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

**Party Responsible for** Section in Protocol for **Laboratory Assessment Performing Test Details** Clinical laboratory tests Central laboratory 9.7.5 Antibody testing BioMarin<sup>a</sup> 9.7.4.2 PK variables **BioMarin** 9.7.3 Blood Phe concentrations Central laboratory 9.7.2.1 Urinalysis, pregnancy test (urine), **Local laboratory** 9.7.5, 9.7.4.1 and sedimentation rate

**Table 9.7.1.1: Summary of Laboratory Assessments** 

## 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, **including allergy history**, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety.

This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

# 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.


Phe, phenylalanine; PK, pharmacokinetic.

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



## 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, weight (kg), and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only.

# 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the final follow-up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

## **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Month 12 and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

# 9.7.2 Efficacy Variable

# 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn in the morning, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 2.1.1).

In addition, after each administration of study drug, the subject will have a blood Phe measurement by fingerstick as outlined in Table 2.1.1. This may be done by the subject at home. Subjects who have their dose frequency increased will have additional Phe assessments performed as outlined in Table 2.1.2 and Table 2.1.3.

A central laboratory will be used for blood Phe concentration analysis.

### 9.7.3 Pharmacokinetic Variables

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (120-600 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks.



Subjects who have increased their dose frequency to twice weekly or daily will have addition PK assessments performed for 5 weeks after the change in dose regimen (refer to Section 12.3.5 and Table 2.1.2 and Table 2.1.3). BioMarin will perform the analysis.

## 9.7.4 Safety Variables

## 9.7.4.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 2.1.1). Female subjects with a positive **serum** pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

# 9.7.4.2 Antibody Testing

Immunogenicity will be assessed by determining antibody response and neutralizing activity with the following measurements: 1) anti-rAvPAL immunoglobulin G (IgG) antibodies, 2) anti-rAvPAL immunoglobulin M (IgM) antibodies, 3) anti-PEG IgG antibodies, 4) anti-PEG IgM antibodies, 5) anti-rAvPAL-PEG immunoglobulin E (IgE) antibodies, and 6) anti-rAvPAL-PEG Enzyme Activity Neutralizing antibodies (NAb). Validated immunogenicity assays will be used per the time points indicated in the Schedule of Events (Table 2.1.1).

BioMarin will perform the analysis except for anti-rAvPAL-PEG IgE antibodies, which will be assessed by a Contract Research Organization.

## 9.7.5 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the result is clinically significant.



The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.

Specific days for obtaining samples are provided in Table 2.1.1 and in Section 12. The scheduled clinical laboratory tests are listed in Table 9.7.5.1. A central laboratory will be used for analysis.



**PAL-003** 


**Table 9.7.5.1: Clinical Laboratory Tests** 

| <b>Blood Chemistry</b> | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if applicable <sup>a</sup> |
| Alkaline<br>Phosphatase | Hematocrit | Color | |
| ALT (SGPT) | WBC count | рН | |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | |
| BUN | Differential cell count | Protein | |
| Creatinine | Sedimentation rate <sup>a</sup> | Glucose | |
| GGT | CRP <sup>b</sup> | Bilirubin | Phenylalanine |
| Total protein | | Nitrite | СН50 <sup>b</sup> |
| Calcium | | Urobilinogen | C <sub>1</sub> b |
| Sodium | | Hemoglobin | C <sub>4</sub> <sup>b</sup> |
| Potassium | | | Serum tryptase level b,c |
| Glucose | | | |
| Uric acid | | | |
| $CO_2$ | | | |
| Chloride | | | |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; **CH50, total hemolytic complement**; CO<sub>2</sub>, carbon dioxide; **CRP, C-reactive protein;** GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.

<sup>&</sup>lt;sup>a</sup> To be performed by local laboratory.

<sup>&</sup>lt;sup>b</sup> Perform for Unscheduled Skin Reaction visit only (within 48 hours of reaction).

<sup>&</sup>lt;sup>c</sup> Perform immediately after reaction if possible.



### 10 REPORTING ADVERSE EVENTS

### 10.1 Adverse Events

According to the ICH definition, an AE (or adverse experience) is "any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the IP."

An adverse drug reaction (ADR) is described by the ICH as "all noxious and unintended responses to a medicinal product related to any dose." This means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility, ie, the relationship cannot be ruled out.

An AE may include intercurrent illnesses or injuries that represent an exacerbation (increase in frequency, severity, or specificity) of pre-existing conditions (eg, worsening of asthma). Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The reporting period for non-serious AEs is the period from the first administration of study drug through the final F/U Visit or at the ETV. If a non-serious AE remains unresolved at the conclusion of the study, the PI and medical monitor will make a joint clinical assessment as to whether continued follow-up of the AE is warranted, and the results of this assessment must be documented. Resolution is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

The Investigator will assess AEs for severity, for relationship to IP, and as to whether the event meets one or more of the definitions of a serious adverse event (SAE; refer to Section 10.2).

The Investigator will determine the severity of each AE and will record it on the source documents and AE CRF, using the CTCAE v 3 grades defined below. Events that are CTCAE grades 4 and 5 are serious events and require completion of both an SAE form and AE eCRF.



| Grade | Description |
|-------|----------------------------------|
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |
| 4 | Life threatening or debilitating |
| 5 | Death related |

The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as "serious," which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the relationship of an AE to the IP and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably<br>Related | The administration of IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE is more likely explained by exposure to the IP than by other factors or causes. |


In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).



**PAL-003** 


#### 10.2 Serious Adverse Events

A SAE is defined as any AE that:

- Results in death.
- Is life threatening, that is, places the subject at immediate risk of death from the event as it occurred. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires in-patient hospitalization or prolongation of an existing in-patient hospitalization. Admission of a subject to the hospital as an in-patient as a result of an AE, even if the subject is released on the same day, qualifies as hospitalization.
- Results in persistent or significant disability or incapacity. An event qualifies as
  resulting in a persistent or significant disability or incapacity if it involves a
  substantial disruption of the subject's ability to carry out usual life functions.
  This definition is not intended to include experiences of relatively minor or temporary
  medical significance.
- Is a congenital anomaly or birth defect, that is, an AE that occurs in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Is an important medical event that does not meet any of the above criteria, but may jeopardize the subject or require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such events are intensive treatment in the emergency room, allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

More than one of the above criteria may apply to any specific event.

The reporting period for SAEs begins earlier than non-serious AEs and is the period from the time of signing of the ICF through 4 weeks after the last dose or at the ETV. SAEs reported to the Investigator outside of this reporting period will be reported to BioMarin if, in good medical judgment, the event has any bearing on the study data. SAEs must be followed by the Investigator until resolution, even if this extends beyond the study-reporting period. Resolution of an SAE is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

Any SAE, whether or not considered related to study drug, will be reported immediately (within 24 hours) to BioMarin Pharmacovigilance by fax using the study-specific SAE Report Form. In addition to the outcome of the SAE, any medication or other therapeutic measures used to treat the event will be recorded on the appropriate CRF page(s). Investigators should not wait to collect additional information that fully documents the event before notifying BioMarin Pharmacovigilance of an SAE. BioMarin may be required to



**PAL-003** 


report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit additional information requested by BioMarin as soon as it becomes available.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

# 10.3 Pregnancy

Pregnancy in a subject or partner should be reported immediately (within 24 hours) to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up Form in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

## 10.4 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the medical monitor any AEs for which the issue of seriousness is unclear or questioned. Contact information for the medical monitor is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:
Fax:
E-mail:




#### 11 APPROPRIATENESS OF MEASUREMENTS

## 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

## 12 STUDY PROCEDURES

## 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

## 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- 12-lead ECG
- Clinical laboratory tests (including hematology, chemistry, and urinalysis)
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in PAL-002, these assessments may be the same used for the **Week 16** Visit of PAL-002, if they occur within 28 days from Day 1.



#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done on the third day following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

## 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs, including weight
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (postdose)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- Predose PK sample
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)



#### 12.3.2 Weekly Visits

The following study activities will be performed at the weekly visits beginning with Week 2:

- Vital signs, including weight
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)
- Predose PK sample
  - O Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.
- Predose blood Phe and plasma tyrosine concentration
  - O Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose plasma Phe and tyrosine assessments may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. The weekly plasma Phe assessment may be replaced with a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes.
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

# 12.3.3 Monthly Visits (Week 4, 8, 12, etc)

## Monthly visits consist of all weekly activities and include additional activities.

The following study activities will be performed at the monthly visits beginning with Week 4:



- Vital signs, including weight
- Clinical laboratory tests
- Chest x-ray (Month 12 visit only)
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)
- Predose PK sample (subjects who are on a stable dosing regimen for ≥3 months only)
  - O Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.
- Predose blood Phe and plasma tyrosine concentration
  - O Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose plasma Phe and tyrosine assessments may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. The weekly plasma Phe assessment may be replaced with a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes.
- Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.



## 12.3.4 Quarterly Visits (Week 12, 24, 36, etc)

Quarterly visits consist of all **weekly and** monthly activities and include additional activities. The following study activities will be performed at the quarterly visits beginning with Week 12:

- Physical examination
- Vital signs, including weight
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)
- Predose PK sample (subjects who are on a stable dosing regimen for ≥3 months only)
  - O Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120-600 μmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.
- Predose blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.



#### 12.3.5 Interim Dosing Visit

Subjects who increase their dose frequency during the study from 1x/week to 2x/week or daily will have additional assessments performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased. If the Interim Dosing Visit coincides with a weekly, monthly, or quarterly scheduled visit, the scheduled visit assessments should also be performed. The following study activities will be performed for the Interim Dosing Visit:

- Vital signs, including weight
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Blood Phe measurement by fingerstick
  - o This may be done by the subject at home.
- PK sample
  - O Subjects increase their dose frequency to 2x/week will have an additional predose PK sample obtained prior to administration of the first 4 doses (ie, for 2 weeks after the dose frequency increase). For the remaining 3 weeks after the dose frequency increase, a PK sample will be obtained weekly prior to the first dose. Refer to Table 2.1.2 for the Interim Dosing Visit schedule.
  - Subjects who have their dose frequency increased to daily will have additional PK samples obtained every day for the first week: 12 hours after the first daily dose and predose every day for the rest of the week. After the first week of daily dosing, subjects will have weekly PK samples obtained for 4 additional weeks. Refer to Table 2.1.3 for the Interim Dosing Visit schedule.

## 12.3.6 Unscheduled Hypersensitivity Reaction Visit

Subjects who have a generalized skin reaction after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 48 hours) the reaction. Subjects who have other systemic symptoms or a large local skin reaction that is not contiguous to the injection site (refer to Section 9.1.1) may have these assessments performed per investigator discretion.

| BIOMARIN | PAL-003 |
|----------|---------|
|----------|---------|

- Injection-site inspection
- Clinical laboratory tests
- Sedimentation rate
- CRP, CH50, C1, and C4
- Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)
- Serum tryptase level
  - o Perform immediately after reaction if possible.
  - Assessment is optional for subjects who have a generalized skin reaction per investigator discretion.
- PK sample
- Assessment of AEs
- Concomitant medications

Subjects should then return to the clinic 4 weeks after their last dose of rAvPAL-PEG for the Early Termination Visit assessments (refer to Section 12.4).



#### 12.4 Early Termination Visit

The Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug.

Subjects who complete an Unscheduled Hypersensitivity Reaction Visit (refer to Section 12.3.6) will be terminated from the study. Subjects will then return 4 weeks after the last dose of study drug for the Early Termination Visit.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)



## 12.5 Final Follow-up Visit

The final follow-up (F/U) Visit will occur 1 week after the final dose of study drug.

The following study activities will be performed at the F/U Visit:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibody, and anti-rAvPAL-PEG IgE)



## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

## 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

Safety will be evaluated on the incidence of AEs, **including serious AEs (SAEs)**, and clinically significant changes in vital signs and laboratory test results.

The verbatim terms reported on CRFs to identify AEs will be coded using MedDRA. Treatment-emergent AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. Changes from baseline in vital signs and laboratory test results will be summarized with descriptive statistics.

# 14.3 Pharmacokinetic Analysis

Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis.

Steady-state PK (predose samples) of rAvPAL-PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentrations (120-600 µmol/L) for a minimum of 2 weeks and no further dose modification is planned.

Should data become available from PAL-002 **that** indicate study drug accumulation should also be measured, additional blood draws **may be added** for PK analysis **as needed but not to exceed 3x/week**.

#### 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.



Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 120-600 µmol/L will be summarized by each scheduled time point.

## 14.5 Determination of Sample Size

Subjects who participated in PAL-002 may be enrolled into this study. No formal sample size calculation was conducted.

## 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.

## 14.7 Interim Analyses

At least one interim analysis may be performed by the sponsor during the study. Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

# 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

| BEOMARIN° PAL-003 |
|-------------------|
|-------------------|

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.



## 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act **independently** in an advisory capacity to BioMarin to monitor **the** safety of rAvPAL-PEG in subjects who participate in the study. Meetings of the DMC can be convened at any time at the discretion of the DMC Chair or the Study Medical Officer. The Chair will be notified by the Study Medical Officer of all SAEs and will receive summaries of other safety data as available. The DMC will review the study data as soon as it is available during the study, on a schedule defined in the DMC Charter, and offer advice on whether or not to proceed, modify or terminate study enrollment on the basis of toxicity. Details regarding the DMC membership and safety data to be reviewed by members will be provided in a charter.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.3.



## 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries. The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment. If the subject has followed the Investigator's instructions, BioMarin will pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures, if these costs are not covered by health insurance or another third party that usually pays these costs. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.



#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent. If an Investigator or institution refuses to allow access to subject records because of confidentiality, arrangements must be made to allow an "interview" style of data verification.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the

| BEOMARIN° PAL-003 |
|-------------------|
|-------------------|

clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.



## 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (eg, subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.



## 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.



**PAL-003** 


## 21 REFERENCES

Armstrong, Hempel, Koling, Chan, Fisher, Meiselman, Garratty. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007.

Chen, Scott. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001.

Davis, Abuchowski, Park, Davis. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981.

Fisch. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000.

Gamez, Wang, Sarkissian, Wendt, Fitzpatrick, Lemontt, Scriver, Stevens. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007.

Ganson, Kelly, Scarlett, Sundy, Hershfield. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006.

Guttler, Azen, Guldberg, Romstad, Hanley, Levy, Matalon, Rouse, Trefz, de la, Koch. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003.

Harris, Chess. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003.

Huttenlocher. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000.

Kaufman. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989.

Koch, Hanley, Levy, Matalon, Matalon, Rouse, Trefz, Guttler, Azen, Platt, Waisbren, Widaman, Ning, Friedman, de la. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003.

Lee, Lilburn, Baudin. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003.



Levy. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003.

Matalon, Surendran, Matalon, Tyring, Quast, Jinga, Ezell, Szucs. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003.

Richter, Akerblom. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983.

Richter, Akerblom. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984.

Rouse, Azen. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004.

Scott, Murad, Koumpouras, Talbot, Eaton. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997.

Scriver CR, Kaufman S. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-709.

Shedlovsky, McDonald, Symula, Dove. Mouse models of human phenylketonuria. Genetics 134[4], 1205-1210. 1993.

Walter, White, Hall, MacDonald, Rylance, Boneh, Francis, Shortland, Schmidt, Vail. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002.

Webster, Didier, Harris, Siegel, Stadler, Tilbury, Smith. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007.



#### 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.



## 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

**Protocol Number: PAL-003** 


I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

| Investigator | Signature | Date |
|---|---|---|
| Printed name: | | |
| accepted for the Sponsor: | | |
| On behalf of BioMarin, I conf<br>bligations as detailed in all a | irm that BioMarin, as a sponsor will co<br>oplicable regulations and guidelines. I value that becomes available during the | will ensure that the PI is |
| obligations as detailed in all ap | oplicable regulations and guidelines. I | will ensure that the PI is |

# **B**OMARIN

#### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Study Title: Long-term Extension of a Phase 2, Open-Label, Dose-

Finding Study to Evaluate the Safety, Efficacy, and

Tolerability of Multiple Subcutaneous Doses of rAvPAL-

PEG in Subjects with PKU

Protocol Number: PAL-003

rAvPAL-PEG (PEGylated recombinant Anabaena **Investigational Product:** 

variabilis phenylalanine ammonia lyase)

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria

BioMarin Pharmaceutical Inc. Sponsor:

> 105 Digital Drive Novato, CA 94949

Development Phase: Phase 2

Sponsor's Responsible

Medical Officer: Clinical Sciences

BioMarin Pharmaceutical Inc.

, MD

105 Digital Drive Novato, CA 94949

Duration: Up to 60 months or until study is terminated

0.001 to a maximum weekly dose of 5.0 mg/kg Dose:

Date of Original Protocol: October 08, 2008 Date of Amendment 1: February 09, 2009 Date of Amendment 2: October 30, 2009 Date of Amendment 3: May 04, 2011


May not be divulged, published, or otherwise disclosed to others without prior written approval

from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.



#### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

**Amendment: 3** 

Date: May 04, 2011

#### RATIONALE AND SUMMARY OF CHANGES

The primary rationale for amending this protocol is to include a substudy to assess the safety, efficacy, pharmacokinetics (PK), and immune response when rAvPAL-PEG treatment is temporarily discontinued and then re-started in subjects.

rAvPAL-PEG is being assessed as a long-term, chronic treatment for patients with PKU, and there is limited safety, efficacy, PK, and immune response information about the effects of a temporary dose interruption. Therefore, a Substudy has been added to this study to explore the effects of stopping and re-starting rAvPAL-PEG treatment. In this Substudy, up to 10 subjects will stop dosing for a period of approximately 4 weeks. During this dosing interruption, subjects will be assessed for safety, efficacy, PK, and immune response and will continue to perform the scheduled study assessments. Subjects are eligible for participation in the Substudy if they are on a stable rAvPAL-PEG dosing regimen (ie, blood Phe levels have been reached at 60-600  $\mu$ mol/L) for 4 weeks in this study, have not reported any serious adverse events (SAEs) during this study, and were not enrolled in Study PAL-004.

Currently, there is no information regarding the PK profile of rAvPAL-PEG when blood Phe levels are at 60-600  $\mu$ mol/L for subjects on a multiple-dose regimen. To address this lack of information, additional PK sampling will be performed prior to the dosing interruption. Upon restarting rAvPAL-PEG, PK sampling will also be performed to allow for collection of drug exposure data (area under the plasma concentration-time curve [AUC] and maximum plasma concentration [C<sub>max</sub>]), absorption rate, and clearance for subjects who have been previously exposed to rAvPAL-PEG in this Substudy. This information will allow for comparisons to be performed with subjects who were naïve to previous rAvPAL-PEG treatment from the Phase 1 study, PAL-001.

Following participation in the Substudy, subjects will return to the rAvPAL-PEG dose level and frequency that they were receiving prior to the dose interruption and will continue participation in the study until completion.

|----------|---------|--------|
|----------|---------|--------|

Because rAvPAL-PEG is a bacterial protein, an immune-mediated reaction and a reduction in efficacy (blood Phe reductions) are possible when rAvPAL-PEG dosing is re-introduced after the dose interruption of the Substudy. However, information from nonclinical studies, antibody results, and safety and efficacy results from the clinical studies to date (JAN2011) have shown that there is no added safety risk or risk of decreased efficacy when rAvPAL-PEG dosing is stopped and then re-started at the same dose level.

- In nonclinical studies using the BTBR Pahenu2 (ENU2) mouse model, an animal model that exhibits characteristics similar to those of PKU patients, a 2-4 week dose-interruption was performed in animals administered 80 mg/kg/week. Following the dose interruption assessment, the animals re-started rAvPAL-PEG dosing at the same dose level (80 mg/kg/week). In this assessment, no safety issues were noted upon re-starting dosing with rAvPAL-PEG and there was an immediate return to stable blood Phe reductions.
- There has not been any immediate immunoglobulin E (IgE)-mediated reactions to rAvPAL-PEG observed following administration of a rAvPAL-PEG injection. All reactions to rAvPAL-PEG have been reported approximately 12-24 hours following administration. To date, 1 out of 33 subjects has tested positive by serology to IgE antibodies without reporting any clinical symptoms to suggest anaphylaxis or a severe systemic reaction. Thus, it is not anticipated that reactions to rAvPAL-PEG are IgE-mediated.
- To date (JAN2011), the clinical experience with re-starting rAvPAL-PEG dosing for subjects from Study PAL-001 who rolled over into Study PAL-002 does not indicate an increased safety risk or a decreased effect on reducing blood Phe levels upon re-introduction of drug.
- Nine subjects who received a single dose of rAvPAL-PEG and completed the Phase 1 study, PAL-001, rolled over into the multiple-dose, Phase 2 study, PAL-002. After a period of several months during which no drug was administered, these 9 subjects restarted rAvPAL-PEG dosing in Study PAL-002 at the same starting doses as was administered in Study PAL-001. There has been no difference to date in the safety profile or efficacy profile of the subjects from Study PAL-001 who rolled over into Study PAL-002 (previously exposed to rAvPAL-PEG) when compared with subjects who were naive to rAvPAL-PEG dosing in Study PAL-002. Although previously exposed subjects had higher and a faster return of anti-PAL and anti-PEG immunoglobulin G (IgG) titers than those of naïve subjects, these results have not been associated with a higher safety risk or efficacy riskbased on information to date.
  - In Study PAL-002, 4 subjects to date have had a protocol-defined (per Protocol Amendment # 3 dated 30APR2010), 2-week washout (no dose



administered) following several weeks of a fixed dose of 0.06 mg/kg/week or 0.1 mg/kg/week rAvPAL-PEG. Following the 2 weeks where no dose was administered, all 4 subjects re-started rAvPAL-PEG dosing at a higher dose with no safety issues reported to date. Blood Phe levels for these 4 subjects have not changed upon re-introduction of dosing.

Clinical experience with subjects who have had to temporarily halt dosing due to an adverse event also provides information that stopping and re-starting rAvPAL-PEG dosing does not appear to increase the risk to subject safety. To date, 10 subjects participating in either PAL-002 or PAL-003 have had to temporarily stop dosing due to an adverse event. All 10 subjects resumed dosing following resolution of the event or per determination by the Investigator that subject safety would not be jeopardized with re-starting dosing. These 10 subjects resumed dosing at a reduced dose level after approximately 1-7 weeks of no dosing. Upon re-starting dosing, none of these 10 subjects have experienced additional safety issues. Eight subjects continue to receive dosing with rAvPAL-PEG (APR 2011) and have subsequently increased their dose level without additional reported adverse events that have resulted in a subsequent dosing interruption.

In summary, because the risk to subject safety and efficacy is expected to be limited upon restarting rAvPAL-PEG, dosing will be re-started at the same dose level for subjects in the Substudy. Re-starting rAvPAL-PEG dosing must be performed in the clinic with post-administration observation performed to monitor subject safety. In addition, subjects will continue to be assessed per the safety assessment and stopping criteria defined in the protocol. Dose decreases for safety and increases also will continue to be performed relative to safety as defined in the protocol. In addition, the Substudy objectives have been added to assess the effect of stopping and re-starting rAvPAL-PEG dosing on safety and tolerability, efficacy (blood Phe concentration), PK, and immune response. The PK analysis has also been revised to accommodate for inclusion of the Substudy.

Additional major changes implemented in this protocol amendment are as follows:

|----------|---------|--------|
|----------|---------|--------|

The maximum allowable rAvPAL-PEG dose of 2.0 mg/kg/week has been increased to 5.0 mg/kg/week to allow for further dose increases. This change is based on available safety and blood Phe information to date (JAN2011) from this ongoing study and from the ongoing Phase 2 study, PAL-002. Experience from this study and Study PAL-002to date (JAN2011) indicates that rAvPAL-PEG administered in doses titrated up to a single administration of 2.0 mg/kg/week does not pose a clinically significant risk to subject safety. The most frequently reported AEs in this study and Study PAL-002 have been nonserious injection-site reactions and headache. The reported injection-site reactions have been self-limited and without sequelae. One SAE (dehydration and urticaria) has been reported to date; the event was reported as not related to treatment with rAvPAL-PEG and resolved. Two days after dosing with rAvPAL-PEG, the subject presented with upper respiratory infection symptoms. The subject was started on for the upper respiratory infection. Twenty-four hours and the third day after dosing with rAvPAL-PEG at 0.1mg/kg, after starting the subject presented with a generalized skin reaction (urticaria). Because the subject had no improvement while on went to the emergency room and was admitted to the hospital for intravenous fluid resuscitation and the stopped. Since this event, this subject has remained in the study and and has continued dosing with rAvPAL-PEG, escalating the dose to 0.6 mg/kg with no additional events reported to date. Despite rAvPAL-PEG being well tolerated in doses up to 2.0 mg/kg/week, many of the subjects in Study PAL-003 have not yet been able to achieve and sustain blood Phe reductions to clinically significant levels (120-600 µmol/L; JAN2011). While some subjects who have been administered 2.0 mg/kg/week rAvPAL-PEG have had > 50% reduction from baseline in blood Phe levels, they have not yet achieved the protocol-defined target blood Phe of 120-600 μmol/L (JAN2011). It is hypothesized that administration of rAvPAL-PEG doses higher than 2.0 mg/kg/week will reduce the blood Phe levels further to within the protocol-defined range of clinical significance (60-600 µmol/L; target range revised per this protocol amendment) without jeopardizing subject safety. Dose increases up to 5.0 mg/kg/week may be implemented if none of the protocol-defined stopping safety criteria are met. Increases to 5.0 mg/kg/week must be performed in increments, every 2 weeks, per the dose increase instructions and safety assessment and stopping criteria outlined for the study. Upwards titration of dose to 5.0 mg/kg/week will be gradual to mitigate risk to subject safety. Also, subjects who increase dosing to up to 5.0 mg/kg/week will continue to be monitored for safety, blood Phe, PK, and antibodies per the scheduled assessments and procedures.

|--------------------------------------|
|--------------------------------------|

- The study inclusion criteria have been modified to permit subjects who have completed Study PAL-004 (A Phase 2, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Dose Levels of rAvPAL-PEG Administered Daily in Subjects with Phenylketonuria) to continue to receive rAvPAL-PEG in this study. Additionally, instruction regarding re-introduction of rAvPAL-PEG dosing has been added for subjects rolling over from Study PAL-004. rAvPAL-PEG treatment will be re-introduced at the same dose level and dosing frequency as was administered at the completion of Study PAL-004. Subjects will be monitored for safety when rAvPAL-PEG dosing is re-started in this study, and subjects will continue to be assessed per the safety assessment and stopping criteria defined in the protocol.
- The target blood Phe level has been revised from 120-600  $\mu$ mol/L to 60-600  $\mu$ mol/L to allow for dosing that may provide greater clinical benefit to subjects. Blood Phe levels of approximately  $60 \pm 13 \ \mu$ mol/L are considered normal per the NIH Consensus Statement, 2000.
- An exploratory objective has been added to assess the relationship of diet and change in blood Phe level in subjects with PKU. Information from a 3-day diet diary will be used to assess dietary Phe intake, as well as all other liquids and food. The study rationale has been revised to include information regarding the relationship of diet in blood Phe concentration following administration of rAvPAL-PEG in subjects with PKU. The study rationale and study outcome measures have also been revised to address this added study objective.
- Information regarding self administration of rAvPAL-PEG has been added. Self-administration of study drug is now allowed by the subject but only if approved by both the Principal Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. This change has been made to increase subject participation and to increase study completion given the long study duration.

Specific revisions to the protocol, including the major changes presented and discussed above, are as follows:

- 1. Information regarding the PAL-003 Substudy has been added.
  - o Substudy objectives have been added for to assess for safety, efficacy, PK, and immune response (refer to the Synopsis [Section 2] and Section 8).
  - The secondary PK objective has been removed; the added PK objective for the Substudy will allow for analysis of PK profile, including clearance, when drug has been stopped and restarted in previously exposed subject who have been administered multiple doses of rAvPAL-PEG (refer to the Synopsis [Section 2] and Section 8), and the PK analysis has been modified to address the Substudy (Section 14.3).



- The Study Rationale has been revised to include information regarding the Substudy (refer to Section 7.3). The nonclinical section (Section 7.1) has also been updated with information regarding nonclinical results relative to stopping and re-starting dosing.
- o Information about the Substudy has been added to the Study Design section (refer to the Synopsis [Section 2] and Section 9.1).
- o Instruction regarding re-starting rAvPAL-PEG dosing following approximately 4 weeks of no dosing has been added (refer to Section 9.1). rAvPAL-PEG dosing will be re-started at the same dose level and dosing frequency as was administered prior to the dosing interruption. The first dose administered following the dose interruption must be performed in the clinic. A follow-up telephone call will be made to monitor subject safety 24 hours following the return to dosing.
- Information regarding the risks of stopping and re-starting rAvPAL-PEG dosing has been added to the Overall Risks and Benefits section (Section 7.4.3).
- Additional PK sampling has been added immediately prior to the dose interruption, during the dose interruption, and for the first week upon restarting rAvPAL-PEG. PK sampling timepoints have been added to Section 9.7.3.
- The Study Procedures (Section 12.3.3) and have been modified to include the Substudy PK sampling, and a Substudy Schedule of Events (Table 2.1.2) has been added.
- 2. The maximum weekly dose amount has been revised from 2.0 mg/kg to 5.0 mg/kg.
  - Information regarding dose increases has been revised; subjects may now increase their dose in increments up to 5.0 mg/kg/week (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, and 4.0 mg/kg/week; refer to the Synopsis [Section 2] and Section 9.1.2.1) provided none of the safety assessment or stopping criteria are met.
  - o Information regarding dose decreases has been revised to include decreases in increments for doses starting at 5.0 mg/kg/week (4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, or 0.001 mg/kg; refer to the Synopsis [Section 2] and Section 9.1.2.2).

|----------|---------|--------|
|----------|---------|--------|

- 3. The target blood Phe level has been revised in this amendment from 120-600 μmol/L to 60-600 μmol/L. All subjects in this study may have their rAvPAL-PEG dose increased to achieve a blood Phe reduction to 60-600 μmol/L (refer to the Synopsis [Section 2], Section 9.1, Section 9.1.2, Section 9.4, Section 9.4.6, Section 9.7.3, Section 14.3, and Section 14.4) provided none of the safety assessment or stopping criteria are met.
  - o Revisions to the criteria for blood Phe level and dosing modifications have been made to align with the target blood Phe level indicated in Study PAL-002 (60-600  $\mu$ mol/L) and Study PAL-004 (  $\leq$  60 $\mu$ mol/L). The individualized rAvPAL-PEG dosing will now be based on reductions in blood Phe level to within a range of 60-600  $\mu$ mol/L. Previously, the individualized rAvPAL-PEG dosing was based on reductions in blood Phe levels to  $\geq$  30% of baseline levels.
- 4. Subjects who have completed Study PAL-004 are now eligible for enrollment into Study PAL-003.
  - The inclusion criterion #1 and exclusion criterion #8 have been revised to allow for inclusion of subjects who have completed Study PAL-004 (refer to the Synopsis [Section 2], Section 9.3.1, and Section 9.3.2).
  - O Instruction regarding re-starting rAvPAL-PEG dosing has been added for subjects who completed Study PAL-004 and who are re-starting rAvPAL-PEG dosing in this study (refer to the Synopsis [Section 2]and Section 9.1) following approximately 4 weeks of no dosing. rAvPAL-PEG dosing will be re-started at the same dose level and frequency as was administered upon completion of PAL-004. A follow-up telephone call will be made to monitor subject safety 24 hours following the return to dosing.
  - o The number of study sites and the number of participating subjects have been increased to accommodate for inclusion of subjects who completed Study PAL-004 (refer to Synopsis [Section 2] and Section 9.1).
- 5. An exploratory objective has been added to assess the long-term effects of diet and change in blood Phe concentration following administration of rAvPAL-PEG (refer to Section 8).
  - Information regarding analysis of diet and change in blood Phe concentration has been added to the Study Rationale (Section 7.3), the Exploratory Efficacy Variable (Section 9.7.4), and the Statistical Analysis (Section 14.4) sections.

- 6. Information regarding diet has been revised. Subjects should no longer modify diet for blood Phe concentrations ≤ 120 μmol/L. Diet should now remain stable during the study unless directed otherwise by the Investigator in consultation with the Sponsor's Medical Officer (refer to Synopsis [Section 2], Section 9.1, and Section 9.6).
- 7. Information regarding the allowed number of missed doses has been added to allow subjects who miss dosing due to reasons other than non-compliance to continue to participate in this long-term extension study. Subjects who miss more than 2 consecutive weekly doses (subjects who are dosed weekly) or 3 consecutive daily doses (subjects who are dosed daily) are allowed to continue in the study (refer to Section 9.4.10). Subjects who miss doses due to subject decision, Sponsor decision, or Investigator decision may continue to participate in this study but must continue to perform the scheduled study assessments for blood Phe levels, pharmacokinetics (PK), antibodies, and safety.
  - o Instructions have been added regarding how to re-start rAvPAL-PEG dosing following a dosing interruption that is not due to subject non-compliance. rAvPAL-PEG dosing will be re-started at the same dose level and frequency as was administered prior to the dosing interruption.
  - O Subjects should continue to perform the scheduled study assessments during any dosing interruption.
- 8. Information regarding the safety assessment criteria (referred to as the stopping criteria in the previous protocol amendment, A2) has been revised to align with the criteria in the other Phase 2 studies, PAL-002 and PAL-004.
  - o The definition of the safety assessment criteria has been revised to better monitor subject safety. Dosing will be halted for subjects who have a Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 event, including a systemic reaction that is assessed by the Investigator as related to treatment with rAvPAL-PEG (Synopsis [Section 2] and Section 9.1.3).
  - The definition of the stopping criteria has been revised to better monitor subject safety. Dosing will be halted for the subjects at the same dose level until a safety evaluation has been completed if 2 or more subjects at a dose level have a Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 event, including a systemic reaction that is assessed by the Investigator as related to treatment with rAvPAL-PEG (Synopsis [Section 2] and Section 9.1.4).


- Subjects who are discontinued from study treatment due to safety will now be asked to remain in the study and to continue to perform the remaining scheduled assessments to continue to collect information, including safety information, until study completion (refer to the Synopsis [Section 2] and Section 9.3.3).
- 9. Based on clinical experience to date (JAN2011) from this ongoing study and ongoing Study PAL-002, reductions in blood Phe to normal levels (ie, 60± 13 μmol/L) have not had clinical consequences to subject safety. Therefore, information regarding the possible toxic effects of low blood Phe has been removed.
  - The Summary of Overall Risks and Benefits (Section 7.4) has been revised; information regarding the possible toxic effects of low blood Phe (Section 7.4.3) has been removed.
- 10. The protocol is being amended to allow for self-administration of rAvPAL-PEG by subjects. This change is to facilitate subject recruitment and subject convenience in this long-term study. Subjects may self administer study drug at home only if the subject meets the protocol-specified requirements, per approval of both the Principal Investigator and the Sponsor's Medical Officer, and if adequate training is demonstrated. Additional information will be provided in the PAL-003 Subject Self-Administration Training Materials (refer to the Synopsis [Section 2] and Section 9.4).
- 11. Information regarding systemic reactions and large local reactions has been revised based on clinical experience from the ongoing Phase 2 study, PAL-002 (refer to Section 9.1.1) and to align with information in the protocols for the other Phase 2 studies, PAL-002 and PAL-004.
  - Subjects who have had a systemic reaction or a large local reaction not contiguous to the injection site during the study are no longer required to discontinue from study treatment. Following the reaction, subjects will temporarily halt treatment and be required to complete the assessments of the Unscheduled Hypersensitivity Reaction visit, including assessment of immunoglobulin E (IgE). Subjects who do not have an IgE-mediated reaction may resume treatment with study drug per the discretion of the Investigator and the Sponsor's Medical Officer with premedication and close monitoring. Subjects who have an IgE-mediated reaction should discontinue from further study treatment but continue to complete the remaining study assessments. Information for including these subjects in this study has been provided in Section 7.4.2.



- An additional assessment to monitor subject safety (ie, a drug-specific immunoglobulin E [IgE] assay) has been developed and validated for use during the study. Subjects who had a systemic reaction in Study PAL-002 or Study PAL-004 must be premedicated with antihistamine and acetaminophen prior to each administration of rAvPAL-PEG in this study (Section 9.1.1.3.3).
- The exclusion criterion (#4) has been revised to allow participation of subjects who have had a previous systemic reaction per the discretion of the Principal Investigator and the Sponsor's Medical Officer (refer to the Synopsis [Section 2] and Section 9.3.2).
- An optional skin biopsy of the affected and not affected area has been added to the Unscheduled Hypersensitivity Reaction Visit for subjects who have had a systemic reaction or a large local reaction not contiguous to the injection site. The biopsy is optional per subject consent and should be taken within 1 week of the reaction (refer to Section 9.1.1.3.3, Section 12.3.7, and Table 2.1.1). The biopsy will allow for further monitoring of subject safety.
- 12. To monitor for subject safety, assessments have been added for subjects who have rAvPAL-PEG dosing administered outside of a scheduled clinic visit, including subjects who are on a daily dosing regimen. AEs, concomitant medications, and an inspection of the injection site will be assessed (refer to Section 12 and Table 2.1.1).
- 13. The safety assessments performed during the Unscheduled Hypersensitivity Reaction visit are now mandatory for subjects who have a systemic reaction or a large local reaction that is not contiguous with the injection site. This revision has been made to align with information in the protocols for the other Phase 2 studies, PAL-002 and PAL-004. Subjects who have been deemed appropriate to continue study treatment must perform the Unscheduled Hypersensitivity Reaction visit assessments prior to resuming dosing with rAvPAL-PEG (refer to Section 9.1.1, Section 12, and Table 2.1.1).
- 14. The secondary objective regarding PK has been removed; rAvPAL-PEG drug exposure will be assessed per the objectives added for the Substudy [Section 2] and Section 8). In addition, the PK assessments for subjects who have reached target Phe levels for at least 2 weeks have been clarified; sampling will be performed once per week for 3 consecutive weeks (refer to Section 9.7.3).
- 15. The Safety Reporting section has been revised for clarity and to align with information in the protocols for the other Phase 2 studies, PAL-002 and PAL-004(refer to Section 10).

|---------------------------------------|
|---------------------------------------|

- 16. The required visits that must be performed in the clinic have been clarified; weekly visits are not required to be performed in the clinic if performed by a home healthcare professional. This change will allow for increased subject compliance (refer to Section 12 and Table 2.1.1).
- 17. The duration of the study has been extended from 24 months to up to 60 months to allow for extended collection of long-term safety information from subjects who are administered rAvPAL-PEG (refer to the Synopsis [Section 2] and Section 9.1).
- 18. The PK assessments have been removed from the Interim Dosing Visit for subjects who increase their dose frequency (refer to Section 12and Table 2.1.3and Table 2.1.4) because PK information will now be obtained from the Substudy.
- 19. Information regarding the timing of dose administration and sampling for PK and blood Phe has been revised; dose administration and sampling no longer need to be performed in the morning but must be performed prior to dose administration. This change has been made to allow for feasibility of dosing for both sites and subjects (refer to Section 9.4.6.1, Section 9.7.2.1, and Section 9.4.6.1).
- 20. Results from the completed Phase 1 study, PAL-001, have been added (Section 7.2.1). Information regarding Phase 2 Study PAL-002 has been updated and information regarding Phase 2 Study PAL-004 has been added to the Background section (refer to Section 7.2).
- 21. Because the systemic allergic skin reactions reported in ongoing Study PAL-002 and this ongoing study to date (JAN2011) have been assessed as variants of delayed allergic reactions and do not typically occur until at least 12-24 hours after dose administration, the immediate post-dose observation period has been reduced. The post-administration observation period has been revised from 2 hours to 30-60 minutes (refer to the Synopsis [Section 2], Section 7.4.2.2, Section 7.4.3, Section 9.1, Section 9.1.1.3.3, Figure 9.1.1.3.1, Section 9.1.2.1, and Section 9.4.10). Subjects who have a systemic reaction regardless of when it occurs relative to dosing are still required to report to the clinic as soon as possible for assessment of safety and to have additional laboratory tests performed (ie, the Unscheduled Hypersensitivity Reaction Visit; refer to Section 12.3.7).
  - Subjects who increase their dosing frequency are no longer required to have the post-administration observation period if the increased frequency does not result in an increase in the total weekly dose amount administered (refer to the Synopsis [Section 2] and Section 9.1.2.1).

| BIOMARIN <sup>®</sup> PAL-003 Page 13 | IN |
|---------------------------------------|----|
|---------------------------------------|----|

- 22. The maximum amount of dose allowed per injection of 1.0 mg/kg has been removed to align with information in the protocols for the other Phase 2 studies, PAL-002 and PAL-004; the dose amount and dosing frequency will be managed per the dose increases and dose decreases outlined per the revised information in this amendment (refer to the Synopsis [Section 2], Section 9.1, and Section 9.1.2).
- 23. Phe (fingerstick) assessments have been added for subjects who modify their dose due to safety. These additional assessments will allow for blood Phe concentration to be assessed more frequently (daily for 3 days) following a change in dose (refer to Synopsis [Section 2], Section 9.1.2.1, and Section 12).
- 24. A chest X-ray has been added to the Screening visit (refer to Section 12 and Table 2.1.1) to monitor for subject safety.
- 25. Nonclinical information has been updated with results from the chronic, repeat-dose studies and updates made to the Investigators Brochure (version 4, 1MAR2011; refer to Section 7.1).
- 26. The Schedule of Events (Table 2.1.1) and the Study Procedure section (Section 12) have been updated to reflect the changes to this amendment.
- 27. Administrative revisions have been made to improve clarity and consistency.

Specific revisions to the text of each section of the protocol (since the protocol amendment finalized on 30OCT2009), including the Synopsis, are outlined in Section 24.



#### 2 SYNOPSIS

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| NAME OF FINISHED PRODUCT: | Page: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |
| phenylalanine ammonia lyase | | |

### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


**STUDY SITES:** Approximately 20 centers in the United States

**PHASE OF DEVELOPMENT:** Phase 2

# **STUDY RATIONALE:**

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding studies (Study PAL-002 and Study PAL-004). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

Because rAvPAL-PEG is being assessed as a long-term chronic treatment for patients with PKU, there is a need to understand the effect of a temporary dosing interruption on the safety, efficacy (blood Phe), PK, and immune response. Therefore, a Substudy has been added to this study to assess the effects of stopping and re-starting rAvPAL-PEG treatment in subjects who are on a variety of rAvPAL-PEG dosing regimens (dose level and frequency). Up to 10 subjects who are on a variety of dosing regimens (dose level and frequency) in this study are eligible for participation in the Substudy and will stop dosing for a period of approximately 4 weeks. During this dosing interruption, subjects will be assessed for safety, efficacy, PK, and immune response and will continue to perform the scheduled study assessments.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary.

#### **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To assess the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

- To assess the safety and tolerability of stopping and re-starting rAvPAL-PEG dosing in a subset of subjects with PKU.
- To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on blood Phe concentration in a subset of subjects with PKU.
- To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on immune response in a subset of subjects with PKU.
- To assess the effect of multiple doses of rAvPAL-PEG on the PK profile, in particular clearance of drug, when drug is stopped in a subset of subjects with PKU who have been previously exposed to rAvPAL-PEG.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### STUDY DESIGN AND PLAN:

This is a long-term extension of the Phase 2, open-label, dose-finding studies, PAL-002 and PAL-004, in approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 5.0 mg/kg/week), provided no dose-limiting toxicity is observed in PAL-002 or PAL-004.

Only subjects who completed the protocol-defined study drug regimen in PAL-002 or PAL-004 will be enrolled into this study. Subjects who enroll from PAL-002 will either continue the dose regimen that was administered upon completion of PAL-002 or start dosing at a higher dose per the dose increase instructions. Subjects who enroll from PAL-002 may start this study at a higher dose level provided there was no interruption in dosing since completion of PAL-002 and enrollment into this study. Subjects who enroll from PAL-004 will re-start rAvPAL-PEG dosing in this study at the same dose level and frequency as was administered upon completion of PAL-004. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing in this study. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigaor in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 and PAL-004 subjects' rAvPAL-PEG dosing will continue in PAL-003. In



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 µmol/L. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The subject has completed the study through the Month 60 visit.
- 4. The study is terminated.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

## PAL-003 Substudy

A subset of up to 10 subjects who are already enrolled and who have consented to participate in this study will be asked to participate in a Substudy to assess the effect that stopping and re-starting treatment with rAvPAL-PEG has on safety, efficacy, PK, and immune response. Subjects will be eligible for participation in the Substudy provided they also meet all of the PAL-003 eligibility criteria, have been on a stable dosing regimen for approximately 4 weeks during this study, have not had any serious adverse events reported during PAL-003, and were not enrolled in Study PAL-004. Subjects participating in the Substudy will have rAvPAL-PEG administration halted for approximately 4 weeks regardless of their dosing regimen (dose level and frequency). rAvPAL-PEG will not be administered during the dose interruption; however, subjects will continue to perform assessments for safety, blood Phe concentration, PK, and immune response. Subjects enrolled into the Substudy will also have additional PK sampling performed prior to the dosing interruption and during the dosing interruption.

|----------|---------|---------|
|----------|---------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

To allow for PK sampling once dosing is stopped, subjects may be admitted to a research facility within 8 hours of stopping dosing where they will reside for at least 24 hours. After the dosing interruption, rAvPAL-PEG administration will be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. Upon re-starting rAvPAL-PEG, the first dose must be administered in the clinic and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Additional PK sampling will also be performed for the first week after the dosing interruption.

#### Dose Modifications:

#### Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

For subjects from PAL-002 only, an individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg)) or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 µmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject.
- The dose may be adjusted by increasing the frequency up to dailyfor a total weekly dose not to exceed 5.0 mg/kg.Subjects who increase their dose frequency will have additional assessments performed (Interim Dosing Visit).
- When a dose is increased, the subject must be observed for 30-60 minutes following the



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.

- Only 1 dose (level or frequency) adjustment is allowed every 2 weeks.
- Blood Phe levels will be measured daily for 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed.

### Dose Decrease Methodology

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe  $(60\text{-}600 \, \mu\text{mol/L})$ , as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for safety (ie, any adverse event that may be improved with a lower, more frequent dose).

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced.

# Safety Assessment Criteria:

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level.

# **Stopping Criteria:**

If 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will be evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### NUMBER OF SUBJECTS PLANNED:

Approximately 100 subjects.

# DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation and all protocol-defined study drug in PAL-002 or PAL-004.
- 2. Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

14 days prior to the administration of study drug.

- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL-002 or PAL-004.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

# INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.  $5 \pm 0.2$  mL to deliver 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with 1.  $5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Upon enrollment into this study, subjects from PAL-002 will be dosed with the same or higher dose than the dose that was administered upon completion of PAL-002. Subjects enrolling from PAL-004, will be administered the same dose that was administered upon completion of PAL-004. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on on available information regarding a subject's blood Phe level (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 6120-600 µmol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses.

## **DURATION OF TREATMENT:**

Up to 60 months.

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

## **CRITERIA FOR EVALUATION:**

Efficacy:

Blood Phe concentrations will be measured.

Immunogenicity:

The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-PEG neutralizing antibodies, and anti-PEG-PAL IgE) will be assessed.

Safety:

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

vital signs, ECG results, X-ray results, and laboratory test results.

Pharmacokinetic:

Plasma concentrations of rAvPAL-PEG will be measured for subjects participating in the Substudy.

## **STATISTICAL METHODS:**

# **Sample Size:**

Subjects who participated in PAL-002 or PAL-004 may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

#### **Safety Analysis:**

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, ECG results, and X-ray results will also be provided.

# **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of



| SUMMARY TABLE | FOR NATIONAL |
|--------------------------|--------------------------------------------------|
| Referring to Part of the | <b>AUTHORITY USE</b> |
| Dossier: | ONLY: |
| Volume: | |
| Page: | |
| Reference: | |
| | Referring to Part of the Dossier: Volume: Page: |

60-600 µmol/L will be summarized by each scheduled time point.

# **Exploratory Analysis:**

For subjects who have received any study drug in this study with any post-treatment blood Phe concentration measurements and diet diary information, the relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will be explored.

# **Substudy Analysis:**

For subjects who completed the Substudy, the effect of stopping and re-starting rAvPAL-PEG dosing on safety, blood Phe level, and immune response will be explored.

# Pharmacokinetic Analysis:

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F).




# 2.1 Schedule of Events

**Table 2.1.1: Schedule of Events** 

| | | Treatment Period <sup>o,c</sup> | | | | Unsched | | |
|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly | Monthly<br>(eg, Wk 4, 8,<br>etc.) | 24, etc.) | Final F/U<br>Visit | Early Term.<br>Visit | Hyper.<br>Reaction<br>Visit.<br>Perform |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at<br>Week 2 | Every 4th week; Perform in addition to weekly procedures | Every 12th week. Perform in addition to monthly procedures | 1 week after<br>final dose | 4 weeks after final dose | within 48 hours; then perform Early Term. procedures |
| Informed consent | X | | | | | | | |
| Medical history, including allergy history, and demographics | X | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | | X | X | X | |
| Vital signs and weight | X | X | X | | | X | X | |
| 12-lead ECG | X | | | | | X | X | |
| Clinical laboratory tests <sup>1</sup> | X | | | X | | X | X | $X^{g}$ |
| Sedimentation rate | | X | | | X | X | X | X |
| Chest x-ray | X | | | X<br>(12-month<br>visit only) | | X | X | |
| Urine pregnancy test <sup>n</sup> | X | X | | X | | X | X | |
| Injection-site inspection <sup>1, k</sup> | | (postdose) | X | | | X | X | X |
| Adverse events <sup>J, K</sup> | Χ← | | | | | >X | X | X |
| Concomitant medications <sup>k</sup> | X | X | X | | | X | X | X |
| Diet query | X | X | X | | | X | X | |
| 3-Day diet diary | | | X | | | X | X | |
| Serum antibodies | | X | | X | | X | X | X |
| Plasma Phe and plasma tyrosine <sup>m</sup> | X | X | X | | | X | X | |
| Plasma Phe (fingerstick)" | | | (3 days<br>postdose) | | | | | |
| Plasma PK sample <sup>o</sup> | | X | X | | | X | X | X |
| Administer IP <sup>p</sup> | | X | X | | | | | |




| | | | Treatme | ent Period <sup>o,c</sup> | | | | Unsched. |
|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly | Monthly<br>(eg, Wk 4, 8,<br>etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Final F/U<br>Visit | Early Term.<br>Visit | Hyper.<br>Reaction<br>Visit.<br>Perform<br>within<br>48 hours; |
| | | | | Every 4th<br>week;<br>Perform in | Every 12th<br>week.<br>Perform in | | | within<br>48 hours;<br>then |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at<br>Week 2 | addition to<br>weekly<br>procedures | addition to<br>monthly<br>procedures | 1 week after<br>final dose | 4 weeks after final dose | perform<br>Early Term.<br>procedures |
| Skin biopsy (optional; affected and not affected area) | | | | | | | | X |
| Serum tryptase level q | | | | | | | | X |

AE, adverse event; C<sub>3</sub>, complement 3; C<sub>4</sub>, complement 4; CH50, total hemolytic complement; CRP, C-reactive protein; D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> It is preferable to perform PAL-003 Screening assessments the same day as PAL-002 Week 16 visit or PAL-004 Week 16 visit so there is no interruption of study drug. If performed on the same day, PAL-002 Week 16 visit or PAL-004 Week 16 visit data may be used. If not, PAL-003 Day 1 must occur ≤ 28 days after PAL-003 Screening.

<sup>&</sup>lt;sup>b</sup> Weekly visits do not require an in-clinic visit if conducted by a home healthcare professional. Monthly visits must be performed in the clinic. Dose modifications must be performed in the clinic. Additional visits may occur if deemed necessary to monitor AEs or blood Phe, adjust dosing etc.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Unscheduled hypersensitivity reaction assessments are mandatory for subjects who have a generalized skin reaction. Subjects who have other systemic symptoms or who have a large local skin reaction that is not contiguous to the injection site may have these assessments performed per investigator discretion. Assessments should be performed within 48 hours of the reaction Subjects who do not have an IgE-mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer with close monitoring. Subjects who remain in the study and continue study treatment must be premedicated. Refer to Section 9.1.1.3.3and Section 12.3.7.

<sup>&</sup>lt;sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.

<sup>&</sup>lt;sup>f</sup> Clinical laboratory tests to include hematology, chemistry, and urinalysis. Refer to Table 9.7.6.1.

<sup>&</sup>lt;sup>g</sup> Subjects who have a systemic reaction or a large local reaction not contiguous with the injection site should be assessed for CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub> within 48 hours of the reaction.

<sup>&</sup>lt;sup>h</sup> If positive or equivocal, perform serum pregnancy test.




<sup>1</sup>It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.

- <sup>n</sup> May be done by the subject at home. Samples should be taken at least 2.5 hours after a meal. Will be performed daily for 3 consecutive days after each dose increase.
- ° The PK blood samples will be collected after the subject has achieved and maintained target blood Phe concentrations (60-600 μmol/L) for a minimum of 2 weeks. Once this target is achieved, once weekly predose PK samples will be collected for 3 consecutive weeks.
- <sup>p</sup> Dosing is up to 5.0 mg/kg/week, including subjects who receive more than 1 dose/week. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency will need to be re-evaluated.
- <sup>q</sup> Mandatory for subjects who have a systemic reaction or a large local skin reaction that is not contiguous to the injection site. Take sample immediately after reaction if possible.

 May 04, 2011

<sup>&</sup>lt;sup>i</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm).

<sup>&</sup>lt;sup>j</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug to the final study visit.

<sup>&</sup>lt;sup>k</sup> Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

<sup>&</sup>lt;sup>m</sup> Samples should be drawn at least 2.5 hours after a meal. If dose is modified by increasing dose level, additional blood Phe concentration testing should be done on the third day following dose adjustment.




**Table 2.1.2: Schedule of Events-Substudy** 

| | | S | ubstudy Period <sup>a</sup> | | |
|---|---|---|---|---|---|
| Substudy<br>Assessments and Events | Final Dose<br>(Day 1) | Day 8 | Day 15 | Day 22 | Re-start Dose<br>(Day 29) |
| Physical examination of | X | X | X | X | X |
| Vital signs and weight | X | X | X | X | X |
| Clinical laboratory tests | X | X | X | X | X |
| Sedimentation rate | X | X | X | X | X |
| Urine pregnancy test <sup>c</sup> | X | X | X | X | X |
| Injection-site inspection <sup>a</sup> | (Pre & postdose) | | | | (postdose) |
| Adverse events | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X |
| Diet query | X | X | X | X | X |
| 3-Day diet diary <sup>e</sup> | X | X | X | X | X |
| Serum antibodies | X | X | X | X | X |
| Plasma Phe and plasma tyrosine | X | (8, 12, and 16 hours/Day 1, 24 hours/Day 2, 48 hours/Day 3, 72 hours/Day 4, 96 hours/Day 5, 144 hours/Day 7, 168 hours/Day 8, 216 hours/Day 10 after Final Dose) | | | (Predose and 24 hours/Day 2, 48<br>hours/Day 3, 72 hours/Day 4, 120<br>hours/Day 6, 168 hours/Day 8 after Re-<br>start Dose |
| Plasma PK sample | (Predose) | (8, 12, and 16 hours/Day 1, 24 hours/Day 2, 48 hours/Day 3, 72 hours/Day 4, 96 hours/Day 5, 144 hours/Day 7, 168 hours/Day 8, 216 hours/Day 10 after Final Dose) | | | X (Predose and 24 hours/Day 2, 48 hours/Day 3, 72 hours/Day 4, 120 hours/Day 6, 168 hours/Day 8 after Restart Dose |
| Administer IP | X | | | | X |

AE, adverse event; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine.

 May 04, 2011

<sup>&</sup>lt;sup>a</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>b</sup> Complete physical examinations to include the evaluation of all major body systems.

<sup>&</sup>lt;sup>c</sup> If positive or equivocal, perform serum pregnancy test.

<sup>&</sup>lt;sup>d</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm).




<sup>e</sup>It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug on Substudy Days 1 and 29. On Substudy Days 8, 15, and 22, it is preferable that the subject complete the diary 3 days immediately prior to the next study visit.

 May 04, 2011




Table 2.1.3: Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to 2x/Week

| | Subjects Who Are Administered rAvPAL-PEG 2x/Week Treatment Period <sup>a, b</sup> | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | First Week After<br>Dose Adjustment | | Second Week After<br>Dose Adjustment | | Third Week After<br>Dose Adjustment | | Fourth Week After<br>Dose Adjustment | | Fifth Week After<br>Dose Adjustment | |
| Assessments and Events | First<br>Dose | Second<br>Dose | First<br>Dose | Second<br>Dose | First<br>Dose | Second<br>Dose | First<br>Dose | Second<br>Dose | First<br>Dose | Second<br>Dose |
| Vital signs and weight | X | X | X | X | X | X | X | X | X | X |
| Injection-site inspection | X | X | X | X | X | X | X | X | X | X |
| Adverse events <sup>c</sup> | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X |
| Blood Phe (fingerstick) <sup>d</sup> | X | X | X | X | X | X | X | X | X | X |

AE, adverse event; D, day; PK, pharmacokinetics; Phe, phenylalanine.

<sup>&</sup>lt;sup>a</sup> The additional Interim Dosing Visit assessments should be performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased to 2x/week. All assessments should be performed predose unless specified otherwise.

<sup>&</sup>lt;sup>b</sup> If the Interim Dosing Visit coincides with a regularly scheduled visit, the scheduled visit assessments should also be performed.

<sup>&</sup>lt;sup>c</sup> If any injection site reaction is observed, the corresponding AE data must specify injection location (identify current vs. previous visit's injection, e.g., right arm vs. left arm).

<sup>&</sup>lt;sup>d</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.




Table 2.1.4: Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to Daily

| | | Subjects Who Are Administered rAvPAL-PEG Daily Treatment Period <sup>a, b</sup> | | | | |
|---|---|---|---|---|---|---|
| | First Day After<br>Dose Adjustment | First Week After<br>Dose Adjustment | Second Week<br>After Dose<br>Adjustment | Third Week After<br>Dose Adjustment | Fourth Week After<br>Dose Adjustment | Fifth Week After<br>Dose Adjustment |
| Assessments and Events | Dose 1 | Doses 2-7 | Doses 8-14 | Doses 15-21 | Doses 22-29 | Doses 30-36 |
| Vital signs and weight | X | X | X | X | X | X |
| Injection-site inspection | X | X | X | X | X | X |
| Adverse events <sup>c</sup> | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X |
| Blood Phe (fingerstick) <sup>d</sup> | X | X | X | X | X | X |

AE, adverse event; D, day; PK, pharmacokinetics; Phe, phenylalanine.

<sup>&</sup>lt;sup>a</sup> The additional Interim Dosing Visit assessments should be performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased to daily. All assessments should be performed predose unless specified otherwise.

<sup>&</sup>lt;sup>b</sup> the Interim Dosing Visit coincides with a regularly scheduled visit, the scheduled visit assessments should also be performed.

<sup>&</sup>lt;sup>c</sup> If any injection site reaction is observed, the corresponding AE data must specify injection location (identify current vs. previous visit's injection, e.g., right arm vs. left arm).

<sup>&</sup>lt;sup>d</sup> May be done by the subject at home. Samples should be taken in the morning, at least 2.5 hours after a meal.




# 3 TABLE OF CONTENTS

| 1 | TIT | LE PAG | E | 1 |
|---|---|---|---|---|
| 2 | SYN | NOPSIS | | 14 |
| | 2.1 | Schedu | ıle of Events | 25 |
| 3 | TAE | BLE OF | CONTENTS | 32 |
| 4 | LIS | T OF AI | BBREVIATIONS AND DEFINITIONS OF TERMS | 36 |
| 5 | ETH | HCS | | 39 |
| | 5.1 | Institut | tional Review Board or Ethics Committee | 39 |
| | 5.2 | Ethical | l Conduct of Study | 39 |
| | 5.3 | Subjec | t Information and Informed Consent | 4( |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 41 |
| 7 | INT | RODUC | CTION | 42 |
| | 7.1 | Noncli | nical Studies | 42 |
| | 7.2 | Previo | us Clinical Studies | 4 |
| | | 7.2.1 | Phase 1 Study PAL-001 | 4 |
| | | 7.2.2 | Phase 2 Studies PAL-002 and PAL-004 | 45 |
| | 7.3 | Study | Rationale | 46 |
| | 7.4 | Summ | ary of Overall Risks and Benefits | 48 |
| | | 7.4.1 | Toxicity Due to Exposure to PEG | 48 |
| | | 7.4.2 | Toxicity Due to an Immunologic Reaction | 49 |
| | | 7.4.3 | Effects of Stopping and Re-Starting rAvPAL-PEG Treatment | 52 |
| 8 | STU | JDY OB | JECTIVES | 55 |
| 9 | INV | ESTIGA | ATIONAL PLAN | 56 |
| | 9.1 | Overal | 1 Study Design and Plan | 56 |
| | | 9.1.1 | Management of Local and Systemic Reactions to rAvPAL-PEG | 58 |
| | | 9.1.2 | Dose Modifications | 63 |
| | | 9.1.3 | Safety Assessment Criteria | 64 |
| | | 9.1.4 | Stopping Criteria | 64 |
| | 9.2 | Discus | sion of Study Design, Including Choice of Control Group | 64 |




| | 9.3 | Calaati | on of Study Population | 65 |
|---|---|---|---|---|
| | 9.3 | | * * | |
| | | 9.3.1 | Inclusion Criteria | |
| | | 9.3.2 | Exclusion Criteria | |
| | | 9.3.3 | Removal of Subjects from Treatment or Assessment | |
| | | 9.3.4 | Subject Identification and Replacement of Subjects | |
| | 9.4 | | ents | |
| | | 9.4.1 | Treatments Administered | |
| | | 9.4.2 | Identity of Investigational Product (IP) | |
| | | 9.4.3 | Storage | 70 |
| | | 9.4.4 | Directions for Administration | 70 |
| | | 9.4.5 | Method of Assigning Subjects to Treatment Groups | 72 |
| | | 9.4.6 | Selection of Doses Used in the Study | 72 |
| | | 9.4.7 | Blinding | 73 |
| | | 9.4.8 | Prior and Concomitant Medications | 73 |
| | | 9.4.9 | Treatment Compliance | 74 |
| | | 9.4.10 | Dose Interruption and Missed Doses | 74 |
| | 9.5 | Investig | gational Product Accountability | 74 |
| | | 9.5.1 | Return and Disposition of Clinical Supplies | 74 |
| | 9.6 | Dietary | or Other Protocol Restrictions | 75 |
| | 9.7 | Efficac | y and Safety Variables | 75 |
| | | 9.7.1 | Efficacy and Safety Measurements Assessed | 75 |
| | | 9.7.2 | Efficacy Variable | 77 |
| | | 9.7.3 | Pharmacokinetic Variables | 77 |
| | | 9.7.4 | Exploratory Efficacy Variable | 77 |
| | | 9.7.5 | Safety Variables | |
| | | 9.7.6 | Clinical Laboratory Assessments | 78 |
| 10 | REP | ORTING | G ADVERSE EVENTS | |
| - | | | e Events | |
| | | | s Adverse Events | |
| | | | ncy | 84 |

| BIO | M | AF | 211 | V |
|-----|---|----|-----|---|
|-----|---|----|-----|---|


| | 10.4 Urgent Safety Measures | 84 |
|----|--------------------------------------------------------------|-----|
| | 10.5 BioMarin Pharmacovigilance Contact Information | |
| 11 | APPROPRIATENESS OF MEASUREMENTS | |
| | 11.1 Safety and Pharmacokinetics | |
| | 11.2 Diet Diary | 87 |
| 12 | STUDY PROCEDURES | |
| | 12.1 Prestudy | 8 |
| | 12.2 Screening Visit | 8 |
| | 12.3 Treatment Period | |
| | 12.3.1 Day 1 (Week 1) | 89 |
| | 12.3.2 Weekly Visits | 90 |
| | 12.3.3 Substudy Visits (Weekly) | 91 |
| | 12.3.4 Monthly Visits (Week 4, 8, 12, etc) | 92 |
| | 12.3.5 Quarterly Visits (Week 12, 24, 36, etc) | 93 |
| | 12.3.6 Interim Dosing Visit | 92 |
| | 12.3.7 Unscheduled Hypersensitivity Reaction Visit | 92 |
| | 12.4 Early Termination Visit | 95 |
| | 12.5 Final Follow-up Visit | 96 |
| 13 | DATA QUALITY ASSURANCE | 97 |
| 14 | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 98 |
| | 14.1 Statistical and Analytical Plans | 98 |
| | 14.2 Safety Analysis | 98 |
| | 14.3 Pharmacokinetic Analysis | 98 |
| | 14.4 Efficacy Analysis | 99 |
| | 14.5 Determination of Sample Size | 99 |
| | 14.6 Handling of Missing Data | 99 |
| | 14.7 Interim Analyses | 99 |
| | 14.8 Changes in the Conduct of the Study or Planned Analyses | 99 |
| 15 | DATA MONITORING COMMITTEE (DMC) | 101 |
| 16 | COMPENSATION, INSURANCE, AND INDEMNITY | 102 |

|---|---|---|
| 17 CASE REPORT FORM | IS AND SOURCE DOCUMENTS | 103 |
| 18 STUDY MONITORING | G AND AUDITING | 105 |
| 19 RETENTION OF REC | ORDS | 106 |
| 20 USE OF INFORMATION | ON AND PUBLICATION | 107 |
| 21 REFERENCES | | 108 |
| 22 INVESTIGATOR RES | PONSIBILITIES | 110 |
| 22.1 Conduct of Study | and Protection of Human Subjects | 110 |
| 24 PROTOCOL AMENDA | MENT TEXT REVISIONS | 112 |
| LIST OF TABLES | | |
| Table 2.1.1: Schedule of E | vents | 25 |
| Table 2.1.2: Interim Dosin | g Schedule, Subjects Whose Dose is In | creased to 2x/Daily28 |
| | g Visit Schedule, Subjects Whose Dose | |
| | g Visit Schedule, Subjects Whose Dose | |
| Table 9.4.4.1: Number of I | njections Required For an Individual V | Veighing 80 kg72 |
| Table 9.7.1.1: Summary of | Laboratory Assessments | 76 |
| Table 9.7.6.1: Clinical Lab | oratory Tests | 79 |
| LIST OF FIGURES | | |




## 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

 $AUC_{0-7 \, days}$  area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen

 $^{\circ}$ C degree Celsius  $C_3$  complement 3  $C_4$  complement 4

CBC complete blood count

CD Compact disk

CFR Code of Federal Regulations
CH50 total hemolytic complement

C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form
CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure
DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up g gram




GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IgE immunoglobulin E
 IgG immunoglobulin G
 IgM immunoglobulin M
 IP investigational product
 IRB Institutional Review Board

IV intravenous kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hgmillimeter of mercuryNAbneutralizing antibodiesNCINational Cancer Institute

NOAEL no observable adverse effect level

OTC over the counter

PAH phenylalanine hydroxylase PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator
PK pharmacokinetics
PKU phenylketonuria

rAvPAL-PEG recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG

RBC red blood cell

SAE serious adverse event SAP Statistical Analysis Plan



SBP systolic blood pressure

SC subcutaneous

SD standard deviation SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase SGPT serum glutamic pyruvate transaminase

US United States
WBC white blood cell

**Definition of Terms:** 

# Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.



## 5 ETHICS

## 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

# 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will



provide written, informed consent before any study-related tests or evaluations are performed.

# 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR Part 50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



# 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Regulatory Affairs Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), urinalysis, and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations. Pharmacokinetic (PK) analysis will be performed by BioMarin.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.



## 7 INTRODUCTION

A comprehensive review of PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

# 7.1 Nonclinical Studies

The nonclinical program for rAvPAL-PEG has characterized the pharmacology, pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC route of administration. Pharmacology was assessed in the BTBR  $Pah^{\rm enu2}$  (ENU2) mouse model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to 2000  $\mu$ M) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to male ENU2 mice, plasma Phe concentrations decreased from approximately 2000  $\mu$ M to < 200  $\mu$ M after 2 dose administrations. An attenuated reduction of blood Phe was seen between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe < 200  $\mu$ M over the entire week, which continued for a total of 15 weeks.

In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a 2-4 week dose interruption and an 11-week dose interruption. Following both dose interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A similar interim attenuated response was observed with the longer dose interruption of approximately 11 weeks. In both of these assessments, no safety issues were noted upon re-starting dosing with rAvPAL-PEG (Lapis, 2007, ASHG 57th Annual Meeting).

Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No respiratory or central nervous system (CNS) effects were seen with SC administration of rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV effects of rAvPAL-PEG administered subcutaneously.

Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats and cynomolgus monkeys. The elimination half-life ( $t_{1/2}$ ) values of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and 44 hours, respectively,

|----------|---------|---------|
|----------|---------|---------|

and exhibited modest area under the plasma concentration-time curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the  $t_{1/2}$  was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum observed plasma concentration ( $C_{max}$ ), along with a long  $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) the AUC and the  $C_{max}$  are roughly linearly proportional.

Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given ≥ 3 mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey.



## 7.2 Previous Clinical Studies

The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU patients who do not respond to treatment with Kuvan<sup>®</sup> or are not compliant with Kuvan<sup>®</sup> treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002 and Study PAL-004) based on data from the completed clinical study, PAL-001, and clinical experience to date (JAN2011) from this ongoing study and the other ongoing Phase 2 study, PAL-002.

# **7.2.1 Phase 1 Study PAL-001**

The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations.

The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 µmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG.

Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows:

- rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg.
- For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level for these 5 subjects was 1113 µmol/L.
- Overall, no clinically significant reductions in blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, 0.01, and 0.03 mg/kg.



For subjects who were administered rAvPAL-PEG at the 3 higher dose levels (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration levels, the calculated PK parameters were a mean T<sub>max</sub> of 89-106 hours, a t<sub>1/2</sub> of 46-120 hours, and an AUC<sub>0-t</sub>, and C<sub>max</sub> that were proportional with dose. Drug exposure was slightly increased with increased dose.

## 7.2.2 Phase 2 Studies PAL-002 and PAL-004

Currently, rAvPAL-PEG is being investigated in two Phase 2 clinical trials (PAL-002 and PAL-004). To date (JAN2011), a total of 33 subjects have been administered rAvPAL-PEG in Study PAL-002 and initiation and recruitment of clinical sites is underway for Study PAL-004.

In PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU), approximately 55 subjects will be enrolled and will be administered multiple doses of rAvPAL-PEG up to 5.0 mg/kg/week. PAL-002 is a 2-part study. In Part 1, subjects will be assigned to 1 of 4 rAvPAL-PEG dose cohorts (0.001, 0.003, 0.01, 0.1 mg/kg, or 1.0 mg/kg). rAvPAL-PEG will be administered at a fixed weekly dose of 0.001 mg/kg (Cohort 1), 0.003 mg/kg (Cohort 2), 0.01 mg/kg (Cohort 3), 1.0 mg/kg (Cohort 4), or 0.1 mg/kg (Part 1 Substudy) for 8 weeks. In Part 2, all subjects who complete Part 1 will be administered an adjustable dose of rAvPAL-PEG for up to an additional 8 weeks. The dose administered in Part 2 may be adjusted by dose level and/or dose frequency to reach a target blood Phe concentration of 60-600 µmol/L. Study PAL-003 (Long-Term Extension of a Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU) is an extension study of PAL-002 and PAL-004. Once subjects have completed Study PAL-002 or PAL-004, they have the option to enroll into PAL-003 and to continue to receive doses of rAvPAL-PEG for up to an additional 60 months.

Study PAL-002 was initiated in September 2009 and is ongoing. The primary objective of this study is to evaluate the effect of multiple doses of rAvPAL-PEG on blood Phe concentrations in subjects with PKU for up to 16 weeks of treatment. The secondary objectives of the study are (1) to evaluate the safety and tolerability of SC injections of multiple dose levels of rAvPAL-PEG, (2) to evaluate the antibody response to rAvPAL-PEG, and (3) to evaluate the PK profile of rAvPAL-PEG in subjects with PKU. The study protocol was amended (30APR2010) to include a substudy of an additional rAvPAL-PEG dose level


(0.1 mg/kg/week) that reduced blood Phe concentrations to clinically significant levels in the Phase 1 study, PAL-001. The protocol was amended again (28MAR2011) to increase the starting dose for Cohort 4 from 0.03 mg/kg/week to 1.0 mg/kg/week. To date (JAN2011), 33 subjects have been enrolled into the study and all 10 subjects of the substudy have been dosed with 0.1 mg/kg rAvPAL-PEG. Additional information about the safety reported to date (JAN2011) is provided in Section 7.4.2.

Study PAL-004 is designed to determine if daily administration of rAvPAL-PEG at daily dose levels (0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day) is safe and effective in reducing and maintaining consistent blood Phe concentrations in subjects with PKU. It is hypothesized that a higher starting dose and frequency will reduce blood Phe concentrations to near-normal levels in a timely manner and will provide the greatest clinical benefit. Considering the concentration and volume of drug that is administered subcutaneously, the only way to increase the rAvPAL-PEG dose is via daily administration. Therefore, in Study PAL-004, a higher starting dose of 0.4 mg/kg will be administered 5 days a week (referred to as daily), a dosing regimen that has been observed to be tolerated and to reduce blood Phe concentrations to clinically meaningful levels in previously exposed subjects in this study. Following completion of Study PAL-004, subjects have the option to enroll into this study and to continue to receive doses of rAvPAL-PEG for up to an additional 60 months.

In this study, subjects in PAL-002 and PAL-004 will continue to be administered the same rAvPAL-PEG that was administered in PAL-002 or PAL-004. If the safety, PK, and blood Phe concentration results from either PAL-002 or PAL-004 indicate that the appropriate level of PEGylation and dosing regimen differs from that administered in PAL-002 or PAL-004, the PEGylation and/or dosing regimen administered in this study may change.

#### 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH. Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003,



Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan<sup>®</sup> is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. rAvPAL-PEG is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits.

Because rAvPAL-PEG is being assessed as a long-term chronic treatment for patients with PKU, there is a need to understand the effect of a temporary dosing interruption on the safety, efficacy (blood Phe), PK, and immune response. To date (JAN2011), there is limited information on the effects of a rAvPAL-PEG dose interruption in subjects with PKU. Therefore, a Substudy has been added to this study to assess the effects of stopping and restarting rAvPAL-PEG treatment in subjects who are on a variety of rAvPAL-PEG dosing regimens (dose level and frequency). Up to 10 subjects who are on a variety of dosing regimens (dose level and frequency) in this study are eligible for participation in the Substudy and will stop dosing for a period of approximately 4 weeks. During this dosing interruption, subjects will be assessed for safety, efficacy, PK, and immune response and will continue to perform the scheduled study assessments. There is no information regarding the pharmacokinetic (PK) profile of rAvPAL-PEG when blood Phe levels are at 60-600 µmol/L for subjects on a multiple-dose regimen. To address this lack of information, additional PK sampling will be performed prior to the dosing interruption. Upon restarting rAvPAL-PEG, PK sampling will also be performed to allow for collection of drug exposure data (area under the plasma concentration-time curve [AUC] and maximum plasma concentration  $[C_{max}]$ , absorption rate, and clearance for subjects who have been previously exposed to rAvPAL-PEG in this Substudy. This information will allow for comparisons to be performed with



subjects who were naïve to previous rAvPAL-PEG treatment from the Phase 1 study, PAL-001.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary.

This study is an extension of the dose-finding studies (PAL-002 and PAL-004). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

## 7.4 Summary of Overall Risks and Benefits

It is not expected that data from PAL-002 or PAL-004 will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

## 7.4.1 Toxicity Due to Exposure to PEG

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg rAvPAL-PEG SC. In rats, both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1).

In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.



#### 7.4.2 Toxicity Due to an Immunologic Reaction

The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylation does not eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing the immunogenicity of the molecule, it is reasonable to expect that some individuals may exhibit immune responses upon exposure to the drug. These immune responses may be clinically irrelevant, cause symptoms of various degrees, or lead to neutralization of biological activity. Subjects participating in clinical trials will be monitored closely with specific antibody titers, sedimentation rates, and complete blood counts (CBCs).

In Study PAL-001, there were 11 subjects (out of 25 subjects in the study) with skin-related reactions (injection-site bruising, erythema, pain, rash, swelling, and urticaria) that occurred following the single administration of rAvPAL-PEG. For all of these subjects, the reactions were generalized skin reactions or injection-site skin reactions that did not compromise other organs and were not life-threatening. These suspected antibody-mediated responses were nonserious and mild or moderate in severity. These subjects are not considered to be at significant risk for antibody-mediated reactions with injection of rAvPAL-PEG during PAL-002, PAL-004, or this study; however, specific precautions for these subjects will be taken during this study to monitor subject safety (refer to Section 9.1.1).

In Study PAL-002, 33 subjects have been dosed to date (JAN2011), including at dose levels of 2.0 mg/kg/week (or 0.4 mg/kg/5 days a week). Most reactions reported in these subjects have been nonserious and mild or moderate in severity. There has been 1 SAE reported to date; the event was reported as not related to treatment with study drug. There have been no reports of anaphylaxis to date (JAN2011). Subjects who have a systemic reaction during this study will undergo a series of assessments to monitor safety, including assessment of IgE antibodies, prior to determining if dosing may resume. Additionally, subjects who have systemic reactions will be premedicated and will be monitored closely for safety (refer to Section 9.1.1.3.3 for additional information regarding continued treatment of subjects with systemic reactions during the study).

|----------|---------|---------|
|----------|---------|---------|

PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.), (Harris, 2003, Nat.Rev.Drug Discov.), however, antibodies against PEG may form when PEG is bound to compounds. (Harris, 2003, Nat.Rev.Drug Discov.), (Richter, 1983, Int.Arch.Allergy Appl.Immunol.). In some instances, development of such antibodies did not result in any significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.) Administration of rAvPAL-PEG may lead to anti-PEG antibody formation, and the duration of this possible effect is not known. This may limit a subject's future ability to be treated with other PEG-containing (eg, Depo-Provera) or PEGylated (eg, PEG-interferon) injectable drugs. It is therefore recommended that any PEG-containing injectable drug administered to subjects after completion of this study be done under medical observation.

## 7.4.2.1 Systemic Skin Reactions

Two out of 25 subjects who were enrolled in Study PAL-001 and received the protocol-defined single dose of rAvPAL-PEG reported systemic skin reactions (generalized skin rash) that were attributed to treatment with study drug. One subject received a single dose of 0.001 mg/kg rAvPAL-PEG, and the other subject received a single dose of 0.01 mg/kg rAvPAL-PEG. One of these events was reported as serious, and the other was reported as nonserious; both events were reported following administration of Depo-Provera injections (medroxyprogesterone injection), an injectable contraception. These allergic reactions are thought to be related to the PEG molecules that are found in both the study drug, rAvPAL-PEG, and Depo-Provera. These reactions are not likely to be experienced concurrent with other birth control medications.

The 2 subjects were administered study drug during PAL-001 and then experienced an allergic reaction following an injection of Depo-Provera. The symptoms of the reactions were hives on the arms and legs and difficulty breathing. The symptoms for both subjects resolved within 1 day following treatment with medication, including the Both subjects were examined by an allergy specialist after they completed participation in PAL-001. A skin prick test with Depo-Provera was administered as part of this examination. One subject had a mild allergic reaction to the test; however, no further reactions or complications were reported following subsequent administration of a full dose of Depo-Provera. Upon study completion, the subject continued to receive regular doses (every 3 months) of Depo-Provera, and no further reactions were reported. The second



subject also had a positive reaction to Depo-Provera following administration of the skin prick test. When a subsequent full dose of Depo-Provera was administered, developed hives, itching, and chills. The subject's symptoms resolved within 1 day of taking medication prescribed by an allergist. See Section 7.2.1 for the results from Study PAL-001.

The active drug substance in rAvPAL-PEG is a bacterial protein that may elicit immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and others. The results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys indicated the formation of anti-rAvPAL antibody titers that did not correspond with observations of injection-site reactions. Quantitation of anti-PEG titers were not assessed in the chronic repeat-dose studies in the rat and monkey. Although results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys did not indicate signs of immune-mediated toxicities, it is possible that the physio-chemical properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG in humans. It is currently unknown whether administration of PEG-containing drugs, such as Depo-Provera, has a sensitizing effect to PEG in rAvPAL-PEG when administered in humans. Because the exact basis for these reported events and their duration is not known, the use of PEG-containing injectable drugs prior to, during, and after this study is prohibited as a precautionary measure (refer to Section 9.3.2 and Section 9.4.8.).

#### 7.4.2.2 Management of Allergic Reactions

Allergic reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 30-60 minutes post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of allergic reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection. Subjects who qualify for self administration of study drug will be provided with emergency resuscitation instructions (refer to Section 9.4 and the Subject Self-Administration Training Materials).

In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for antibody testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of allergic symptoms:



- Maintain the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. Acetaminophen or ibuprofen (5-10 mg/kg) may also be administered. An allergy and/or immunology consultation should be sought if necessary. Information regarding the management of local skin, large local skin, and systemic reactions is provided in Section 9.1.1. Detailed instructions for the management of allergic reactions are provided in the Study Reference Manual.

# 7.4.3 Effects of Stopping and Re-Starting rAvPAL-PEG Treatment

The effects of starting, stopping, and re-starting rAvPAL-PEG dosing on safety and blood Phe reductions previously achieved through rAvPAL-PEG dosing are not well defined, and there is limited clinical experience with rAvPAL-PEG. Allergic reactions are a common and expected clinical outcome of re-starting biologic drugs, such as rAvPAL-PEG, and may occur when subjects re-start rAvPAL-PEG dosing. However, no information reported from the ongoing clinical studies, including this study, or nonclinical results point to an increased safety risk or decreased efficacywhen rAvPAL-PEG dosing is stopped and then re-started at the same dose level.

• Nonclinical experience in the BTBR *Pah*<sup>enu2</sup> (ENU2) mouse model indicates that dosing interruptions of 2-4 weeks for mice administered rAvPAL-PEG 80 mg/kg/week had no increased safety risk upon re-starting dosing and there was an immediate return to stable blood Phe reductions (refer to Section 7.1).



PAL-003


- Antibody results from the ongoing Phase 2 study, PAL-002, and this ongoing study to date (JAN2011) have not indicated an immune response that points to an increased safety risk or decreased efficacy upon re-introduction of drug. There has not been any immediate immunoglobulin E (IgE)-mediated reactions to rAvPAL-PEG observed following administration of a rAvPAL-PEG injection. All reactions to rAvPAL-PEG have been reported approximately 12-24 hours following administration. To date, 1 out of 33 subjects has tested positive by serology to IgE antibodies without reporting any clinical symptoms to suggest anaphylaxis or a severe systemic reaction. Thus, it is not anticipated that reactions to rAvPAL-PEG are IgE-mediated.
- To date (JAN2011), the clinical experience with re-starting rAvPAL-PEG dosing for subjects from Study PAL-001 who rolled over into Study PAL-002 does not indicate an increased safety risk or a decreased effect on reducing blood Phe levels upon re-introduction of drug.
  - Nine subjects who received a single dose of rAvPAL-PEG and completed the Phase 1 study, PAL-001, rolled over into the multiple-dose, Phase 2 study, PAL-002. After a period of several months during which no drug was administered, these 9 subjects re-started rAvPAL-PEG dosing in Study PAL-002 at the same starting doses as was administered in Study PAL-001. There has been no difference to date in the safety profile or efficacy profile of the subjects from Study PAL-001 who rolled over into Study PAL-002 (previously exposed to rAvPAL-PEG) when compared with subjects who were naive to rAvPAL-PEG dosing in Study PAL-002. Although previously exposed subjects had higher and a faster return of anti-PAL and anti-PEG IgG titers than those of naïve subjects, these results have not been associated with a higher safety risk or efficacy riskbased on information to date.
  - o In Study PAL-002, 4 subjects to date have had a protocol-defined (per Protocol Amendment # 3 dated 30APR2010), 2-week washout (no dose administered) following several weeks of a fixed dose of 0.06 mg/kg/week or 0.1 mg/kg/week rAvPAL-PEG. Following the 2 weeks where no dose was administered, all 4 subjects re-started rAvPAL-PEG dosing at a higher dose with no safety issues reported to date. Blood Phe levels for these 4 subjects have not changed upon re-introduction of dosing.
  - Clinical experience with subjects who have had to temporarily halt dosing due to an adverse event also provides information that stopping and re-starting rAvPAL-PEG dosing does not appear to increase the risk to subject safety. To date, 10 subjects participating in either PAL-002 or PAL-003 have had to

|----------|---------|---------|
|----------|---------|---------|

temporarily stop dosing due to an adverse event. All 10 subjects resumed dosing following resolution of the event or per determination by the Investigator that subject safety would not be jeopardized with re-starting dosing. These 10 subjects resumed dosing at a reduced dose level after approximately 1-7 weeks of no dosing. Upon re-starting dosing, none of these 10 subjects have experienced additional safety issues. Eight subjects continue to receive dosing with rAvPAL-PEG (APR 2011) and have subsequently increased their dose level without additional reported adverse events that have resulted in a subsequent dosing interruption.

In this study, measures will be taken to reduce the risk to subject safety upon re-starting rAvPAL-PEG dosing while still allowing for reductions in blood Phe level to clinical significance (blood Phe reduction to 60-600 µmol/L). To mitigate the possible safety risks upon re-starting rAvPAL-PEG dosing, re-introduction of dosing should be performed in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call should be made to subjects 24 hours following re-starting of dosing to monitor subject safety. Subjects will also continue to be assessed per the safety assessment and stopping criteria defined in Section 9.1.3 and Section 9.1.4, and dose decreases will continue to be performed relative to safety as defined in Section 9.1.2.2. To mitigate the possible reduced effect on blood Phe level upon re-starting rAvPAL-PEG, subjects in this study who interrupt dosing whether per the protocol (ie, subjects participating in the Substudy; refer to Section 9.1) or for other reasons (refer to Section 9.4.10) will re-start rAvPAL-PEG dosing at the same dose level.



#### 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To assess the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

- To assess the safety and tolerability of stopping and re-starting rAvPAL-PEG dosing in a subset of subjects with PKU.
- To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on blood Phe concentration in a subset of subjects with PKU.
- To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on immune response in a subset of subjects with PKU.
- To assess the effect of multiple doses of rAvPAL-PEG on the PK profile, in particular clearance of drug, when drug is stopped in a subset of subjects with PKU who have been previously exposed to rAvPAL-PEG.



#### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of the Phase 2, open-label, dose-finding studies, PAL-002 and PAL-004, in approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 5.0 mg/kg/week), provided no dose-limiting toxicity was observed in PAL-002 or PAL-004.

Only subjects who completed the protocol-defined study drug regimen in PAL-002 or PAL-004 will be enrolled into this study. Subjects who enroll from PAL-002 will either continue the dose regimen that was administered upon completion of PAL-002 or start dosing at a higher dose per the dose increase instructions. Subjects who enroll from PAL-002 may start this study at a higher dose level provided there was no interruption in dosing since completion of PAL-002 and enrollment into this study. Subjects who enroll from PAL-004 will re-start rAvPAL-PEG dosing in this study at the same dose level and frequency as was administered upon completion of PAL-004. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing in this study. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to each clinic visit for review with the clinical study staff.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self administration. Additional information is provided in the Subject Self-Administration Training Materials.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.



In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 and PAL-004 subjects' rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 µmol/L. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 2.1.1, Table 2.1.2, Table 2.1.3 and Table 2.1.4 (Schedule of Events). After the subject's blood Phe concentration has been controlled to within a target range (60-600 μmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

A subject will continue in PAL-003 until one of the following occurs:

- 1. The subject withdraws consent and discontinues from the study.
- 2. The subject is discontinued from the study at the discretion of the Investigator.
- 3. The subject has completed the study through the Month 60 visit.
- 4. The study is terminated.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

A subset of up to 10 subjects who are already enrolled and who have consented to participate in this study will be asked to participate in a Substudy to assess the effect that stopping and re-starting treatment with rAvPAL-PEG has on safety, efficacy, PK, and immune response. Subjects will be eligible for participation in the Substudy provided they also meet all of the PAL-003 eligibility criteria, have been on a stable dosing regimen for approximately 4 weeks during this study, have not had any serious adverse events reported during PAL-003, and were not enrolled in Study PAL-004. Subjects participating in the Substudy will have rAvPAL-PEG administration halted for approximately 4 weeks regardless of their dosing regimen (dose level and frequency). rAvPAL-PEG will not be administered during the dose



interruption; however, subjects will continue to perform assessments for safety, blood Phe concentration, PK, and immune response. Subjects enrolled into the Substudy will also have additional PK sampling performed prior to the dosing interruption and during the dosing interruption. To allow for PK sampling once dosing is stopped, subjects may be admitted to a research facility within 8 hours of stopping dosing where they will reside for at least 24 hours. After the dosing interruption, rAvPAL-PEG administration will be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. Upon re-starting rAvPAL-PEG, the first dose must be administered in the clinic and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Additional PK sampling will also be performed for the first week after the dosing interruption.

## 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEG

Subjects who qualify for self administration of study drug will be provided with information and instruction with regard to management of local and systemic reactions (refer to the Subject Self-Administration Training Materials).

# 9.1.1.1 Subjects Who Have Had Previous Hypersensitivity Reactions to rAvPAL-PEG or a PEG-containing Product

Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from PAL-002 or PAL-004 are excluded from participation in this study. Subjects who experienced a generalized skin rash are included in this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in PAL-002 or PAL-004 are eligible to participate in this study. Subjects who have had a previous reaction and are deemed eligible for participation must be premedicated orally with acetaminophen and/or antihistamines 1 hour prior to study drug dosing for the remainder of the study. The premedication dosage will be standard. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). Subjects may develop systemic, large local skin, or local skin reactions after enrollment in PAL-003. Refer to Section 9.1.1.2 for definitions of systemic and local skin reactions. For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.



# 9.1.1.2 Definition of Hypersensitivity Reactions to rAvPAL-PEG Administered Subcutaneously

During Study PAL-003, subjects may experience hypersensitivity reactions to rAvPAL-PEG. The hypersensitivity reactions are defined as follows:

#### Local skin reaction:

- Skin signs or symptoms in 1 affected primary location, ie, hives, wheals, or swelling or an area of erythema, redness, induration, pain, or itching at or near the site of injection.
- Large local skin reaction:
- Skin signs or symptoms, ie, hives, wheals, or swelling or an area of erythema, redness, or induration with pain or itching that extends beyond the site of injection by approximately 6 inches (15 cm) and/or signs or symptoms that are not contiguous to the injection site. These may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure and, therefore, will be managed as a systemic reaction when not contiguous to the injection site.
- Systemic reaction (including generalized skin symptoms):
- Skin and non-skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological; and/or a fever attributed to treatment with rAvPAL-PEG (≥ 100.4°F or ≥ 38°C).

For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.



|----------|---------|---------|
|----------|---------|---------|



 May 04, 2011



#### 9.1.1.3.1 Local Skin Reactions

Subjects who have had a local skin reaction (refer to Section 9.1.1.2 for definition) after administration of rAvPAL-PEG in this study may continue if the symptoms do not worsen and no other symptoms have developed but may be premedicated with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to the next dose of study drug dosing. Because antihistamines can cause drowsiness, it should be administered only if the subject is accompanied by a designated driver.

Symptoms of local reactions may be treated with local application of ice and non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.2.2).

If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from study treatment.

#### 9.1.1.3.2 Large Local Skin Reactions

Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be contiguous to the rAvPAL-PEG injection site, and subjects with either type of large local skin reaction may continue dosing if the skin symptoms have resolved and no other symptoms have developed. Subjects may be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing.

#### 9.1.1.3.2.1 Large Local Skin Reactions Contiguous to Injection Site

Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may remain in the study if the skin symptoms have resolved and no other symptoms have developed. For the remainder of the study, subjects may be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to the next dose of study drug. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable).

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

#### 9.1.1.3.2.2 Large Local Skin Reactions Not Contiguous to Injection Site

Large local skin reactions that are not contiguous to the injection site may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure to rAvPAL-PEG and, therefore, will be managed as a systemic reaction (refer to Section 9.1.1.3.3). An example of



a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk.

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

#### 9.1.1.3.3 Systemic Reactions

Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a definition) after administration of rAvPAL-PEG must stop further administrations of rAvPAL-PEG and must immediately return to the clinic for safety assessments . Subjects who experience generalized skin symptoms are included in this category. Immediately after the systemic reaction (within 48 hours), subjects with generalized skin symptoms must have additional assessments performed for safety (ie, Unscheduled Hypersensitivity Reaction Visit): serum antibodies (anti--PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, anti-rAvPAL-PEG neutralizing antibodies); serum tryptase level (it is recommended that this sample be drawn immediately after reaction); sedimentation rate; CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub>; skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction); and clinical laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1).

Following completion of the Unscheduled Systemic Reaction Visit, administration of rAvPAL-PEG may resume up to 1 week following the onset of the reaction if the systemic reaction is not IgE-mediated and the subject's safety will not be further compromised with resumed dosing. rAvPAL-PEG administration will resume at the next lowest dose level. Restarting of rAvPAL-PEG administration following a systemic reaction must be performed in the clinic for the first week of resumed dosing. Subjects must be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing for the remainder of the study. Additionally, subjects must be closely monitored for 30-60 minutes following every administration of study drug. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

If blood Phe concentrations are not 60-600  $\mu$ mol/L following 1 week of daily administration at the lowered dose cohort and there is no further evidence of toxicity (ie, another systemic reaction attributed to rAvPAL-PEG administration or clinically significant abnormal laboratory test results), the subject may be administered the next highest dose level in the clinic per the allowable dose increases outlined in Section 9.1.2. Subjects must be



premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing for the remainder of the study. Additionally, subjects must be closely monitored for 30-60 minutes following every study drug administration. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

#### 9.1.2 Dose Modifications

# 9.1.2.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

For subjects from PAL-002, an individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg) or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject.
- The dose may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 5.0 mg/kg.Subjects who increase their dose frequency should perform the Interim Dosing Visit assessments (refer to Section 12.3.6 and Table 2.1.3 and Table 2.1.4).
- When a dose is increased, the subject must be observed for 30-60 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose (level or frequency) adjustment is allowed every 2 weeks.
- Blood Phe levels will be measured daily for 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed.



#### 9.1.2.2 Dose Decrease Methodology

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse event (any hypersensitivity reaction as defined in Section 9.1.1.2). Dose decreases may occur for safety (ie, any adverse event that may be improved with a lower, more frequent dose).

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced.

### 9.1.3 Safety Assessment Criteria

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principle Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level.

## 9.1.4 Stopping Criteria

If 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate.

# 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.



#### 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation and all protocol-defined study drug in PAL-002 or PAL-004.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

#### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.



- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination fro PAL-002 or PAL-004.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

## 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study treatment should continue to perform the study tests and evaluations until study completion. For subjects who discontinue from the study, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study treatment include, but are not limited to, the following:



- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.

If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

#### 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in PAL-002 or PAL-004. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.



#### 9.4 Treatments

Upon enrollment into this study, subjects from PAL-002 will be dosed with the same or higher dose that was administered upon completion of PAL-002. Subjects enrolling from PAL-004, will be administered the same dose that was administered upon completion of PAL-004. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed to by the PI and the Study Medical Officer, based upon the subject's response to doses.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects may be eligible to self administer study drug if he or she meets the following criteria:

- The subject is on a stable dosing regimen for 2 weeks.
- The subject has not experienced any CTCAE Grade 3 or higher adverse event.
- The subject has not experienced any hypersensitivity reaction to rAvPAL-PEG for at least 4 weeks.
- The subject has no cognitive impairments that may increase the safety risk of self administration per the assessment of the PI.
- The subject has been approved for self administration of study drug by the Sponsor's Medical Officer.
- The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely.
- The subject has been provided with epinephrine and has been trained on when and how to administer it.

Qualified study site personnel will train each eligible subject on all procedures for self administration of study drug under the supervision of the PI. Qualified study site personnel will also be required to observe the subject prepare and perform at least 1 injection prior to allowing the subject to self administer a dose at home. The patient will see a study site nurse



or home healthcare nurse in person every week to ensure that the subject continues to perform all self-administration procedures correctly, to assess of adverse events, and to answer questions throughout the duration of the study. The study site nurse or home healthcare nurse will also perform the regularly scheduled assessments and procedures as outlined in Table 2.1.1 and Section 12; the subject must perform a clinic visit monthly at minimum. Training materials and other information specific to the study site personnel are provided in the Subject Self-Administration Training Materials.

Subjects who are eligible for self administration will be provided with a Subject Study Manual. Self-administration training materials will be provided in the Subject Study Manual to supplement the in-person training provided by the qualified study site personnel. The Subject Study Manual will include step-by-step instruction on the following:

- How to prepare and perform the injections of study drug safely.
- How to receive, track, store, prepare, and return both used and unused study drug.
- How to safely use and dispose of syringes used for injections of study drug.
- How to use a new syringe and vial every time drug is administered.
- How to care for their injection site after an injection of study drug.
- How to identify an adverse reaction and how to report this reaction to the study site.
- How and when to use epinephrine.
- Who to contact at the study site in case of an emergency.

The PI or the Sponsor's Medical Officer may request that self administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse.

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site or subject with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplying the study drug to subjects who qualify for self administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites.

Information regarding supplying study drug to subjects who qualify for self administration is provided in the Subject Self-Administration Training Materials.



## 9.4.2 Identity of Investigational Product (IP)

#### 9.4.2.1 Product Characteristics and Labeling

The rAvPAL-PEG drug product for SC injection is formulated and supplied as a sterile aqueous (colorless to pale yellow) solution in clear, single-use, type-1 borosilicate glass vials. Each 3 mL vial contains  $1.5 \pm 0.2$  mL to deliver 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with  $1.5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Dilution instructions are provided in a separate instruction manual.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

Drug product packaging will be identified with the lot number and expiration date, and will be provided in a box labeled with the study number.

## 9.4.3 Storage

IP must be stored at  $5 \pm 3$  °C ( $41 \pm 5$  °F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

Specific instructions for storage of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg.

Dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

|----------|---------|---------|
|----------|---------|---------|

The injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). The number of injections required for an individual weighing 80 kg (about 176 pounds) is provided in Table 9.4.4.1 as an example. Note this table is for example purposes only. Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff or other qualified and trained study personnel.

Information for subjects who are participating in the Substudy and re-start rAvPAL-PEG dosing is provided in Section 9.1. Information for dosing of subjects who enroll into this study after completing Study PAL-004 is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10.

Instructions for administration of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials.



Table 9.4.4.1: Number of Injections Required For an Individual Weighing 80 kg

| Dose Group<br>(mg/kg) | Weight (kg) | Volume of Study Drug<br>(mL) <sup>a</sup> | No. of<br>Injections <sup>b</sup> |
|---|---|---|---|
| 0.001 | 80 | 0.8 | 1 |
| 0.003 | 80 | 0.6 | 1 |
| 0.01 | 80 | 0.8 | 1 |
| 0.03 | 80 | 0.2 | 1 |
| 0.06 | 80 | 0.5 | 1 |
| 0.1 | 80 | 0.8 | 1 |
| 0.3 | 80 | 2.4 | 2 |
| 0.6 | 80 | 4.8 | 2 or 3 |
| 1.0 | 80 | 8.0 | 4 |

aStudy drug is supplied at a concentration of 10 mg/mL and is then diluted by differential amounts as specified in the PAL-003 Pharmacy Manual. Volume to be injected is calculated based on a starting volume.

Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may need to be re-evaluated (refer to Section 9.4.10).

# 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in PAL-002 or PAL-004.

#### 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study and the ongoing study, PAL-002, to date (JAN2011).

<sup>&</sup>lt;sup>b</sup>Number of injections per dose is dependent upon site policy for SC injections. The number of injections may vary at the discretion of the Investigator.



#### 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered by clinic staff or other qualified and trained study personnel.

Subjects may self administer study drug at home if approved by the Sponsor's Medical Officer and if adequate training is provided (refer to Section 9.4).

## 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the medical monitor must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in PAL-002 or PAL-004) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior local skin reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and/or antihistamines (refer to Section 9.1.1). If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior systemic reaction to rAvPAL-PEG or a PEG-containing product may participate in this study (refer to Section 9.1.1).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.



#### 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

# 9.4.10 Dose Interruption and Missed Doses

Information for subjects who are participating in the Substudy and re-start rAvPAL-PEG dosing is provided in Section 9.1. Information for dosing of subjects who enroll into this study after completing Study PAL-002 or Study PAL-004 is provided in Section 9.1.

During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator in consultation with the Sponsor's Medical Officer. Subjects who miss more than 2 consecutive weekly doses (weekly dosing schedule) or 3 consecutive daily doses (daily dosing schedule) for whatever reason may continue participation in this study. After a dosing interruption, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects should continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 2.1.1, Table 2.1.2, Table 2.1.3 and Table 2.1.4) during any dosing interruption.

Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study treatment per discretion of the Sponsor or Investigator (refer to Section 9.3.3).

#### 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), IP returned, and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

### 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.



Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

Subjects who qualify for self administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials).

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

## 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigaor in consultation with the Sponsor's Medical Officer.

A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next dose of study drug. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4.

### 9.7 Efficacy and Safety Variables

## 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis (Section 2.1) describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.



**Table 9.7.1.1: Summary of Laboratory Assessments** 

| Laboratory Assessment | Party Responsible for<br>Performing Test | Section in Protocol for Details |
|---|---|---|
| Clinical laboratory tests | Central laboratory | 9.7.6 |
| Antibody testing | BioMarin <sup>a</sup> | 9.7.5.2 |
| PK variables | BioMarin | 9.7.3 |
| Blood Phe concentrations | Central laboratory | 9.7.2.1 |
| Urinalysis, pregnancy test (urine), and sedimentation rate | Local laboratory | 9.7.6, 9.7.5.1 |

Phe, phenylalanine; PK, pharmacokinetic.

## 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, including allergy history, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

#### 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

# 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, weight (kg), and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only.

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



## 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the Final Follow-Up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

# **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Screening, Month 12, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

# 9.7.2 Efficacy Variable

## 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 2.1.1, Table 2.1.2, Table 2.1.3 and Table 2.1.4).

In addition, after each administration of study drug, the subject will have a blood Phe measurement by fingerstick as outlined in Table 2.1.1, Table 2.1.2, Table 2.1.3 and Table 2.1.4. This may be done by the subject at home.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Subjects enrolled in the Substudy will have additional PK sampling performed prior to the planned dosing interruption and upon re-introduction of rAvPAL-PEG. For subjects participating in the Substudy, PK sampling will be performed as follows:

- When dosing is stopped, PK sampling will be performed prior to the final dose and then postdose at 8 hours, 12 hours, 16 hours, 24 hours, 48, hours, 72 hours, 96 hours, 144 hours, 168 hours, and 216 hours.
- When dosing is re-started, PK sampling will be performed predose and then postdose at 24 hours, 48 hours, 72 hours, 120 hours, and 168 hours.

BioMarin will perform the anlaysis.

## 9.7.4 Exploratory Efficacy Variable

Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits. Subjects will be instructed to record all



food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each week. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator.

# 9.7.5 Safety Variables

# 9.7.5.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 2.1.1 and Table 2.1.2). Female subjects with a positive serum pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

# 9.7.5.2 Antibody Testing

Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgE, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1.3.3). Validated immunogenicity assays will be used per the time points indicated in the Schedule of Events (Table 2.1.1 and Table 2.1.2).

BioMarin will perform the analysis except for IgE antibodies, which will be assessed by a Contract Research Organization.

#### 9.7.6 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not any abnormal result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.

|-----------------------|---------|---------|
|-----------------------|---------|---------|

Specific days for obtaining samples are provided in Table 2.1.1, Table 2.1.2, and in Section 12. The scheduled clinical laboratory tests are listed in Table 9.7.6.1. A central laboratory will be used for analysis.

**Table 9.7.6.1: Clinical Laboratory Tests** 

| Blood Chemistry | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if applicable <sup>a</sup> |
| Alkaline<br>Phosphatase | Hematocrit | Color | |
| ALT (SGPT) | WBC count | pН | |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | |
| BUN | Differential cell count | Protein | |
| Creatinine | | Glucose | |
| GGT | | Bilirubin | Phenylalanine |
| Total protein | | Nitrite | CH50 <sup>b</sup> |
| Calcium | | Urobilinogen | $C_1^{b}$ |
| Sodium | | Hemoglobin | C <sub>4</sub> <sup>b</sup> |
| Potassium | | | $C_3^b$ |
| Glucose | | | Serum tryptase level b,c |
| Uric acid | | | Sedimentation rate <sup>a</sup> |
| $CO_2$ | | | CRP <sup>b</sup> |
| Chloride | | | |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; C, complement; CH50, total hemolytic complement; CO2, carbon dioxide; CRP, C-reactive protein; GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.

<sup>&</sup>lt;sup>a</sup> To be performed by local laboratory. If urine pregnancy test is positive or equivocal, serum sample will be taken and assessed by a central laboratory.

<sup>&</sup>lt;sup>b</sup> Perform for Unscheduled Hypersensitivity Reaction visit only (within 48 hours of reaction).

<sup>&</sup>lt;sup>c</sup> Perform immediately after reaction if possible.



#### 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a patient administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment runin).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The study period during which all non-serious AEs and SAEs will be reported begins after informed consent is obtained and the first administration of study drug and continues until 4 weeks following the last administration of study drug or the last visit of the treatment period (refer to Section 12). After informed consent but prior to initiation of study treatment, only SAEs associated with any protocol-imposed interventions will be reported. The criteria for determining, and the reporting of SAEs is provided in Section 10.2.

The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or study participation is not the cause of the AE. Resolution of AEs (with dates) should be documented on the appropriate CRF page(s) and in the subject's medical record.

The Investigator responsible for the care of the subject or qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to seriousness, which is based on patient/event outcome or action criteria usually associated



with events that pose a threat to a patient's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the severity of each AE using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.

| Grade | Description |
|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life-<br>threatening: hospitalization or prolongation of hospitalization<br>indicated; disabling; limiting self care activities of daily<br>living (ADL) |
| 4 | Life threatening or debilitating: consequences; urgent intervention indicated <sup>b</sup> |
| 5 | Death related to AE |

Grade 4 and 5 AEs should always be reported as SAEs.

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

<sup>&</sup>lt;sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.
| BIOMARIN <sup>®</sup> PAL-003 Page 82 | BIOMARIN | PAL-003 | Page 82 |
|---------------------------------------|----------|---------|---------|
|---------------------------------------|----------|---------|---------|

The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time AND The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably<br>Related | The administration of IP and the occurrence of the AE are reasonably related in time AND The AE is more likely explained by exposure to the IP than by other factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).



#### 10.2 Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Is fatal.
- Is life threatening.
- Note: Life-threatening refers to an event that places the patient at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires or prolongs inpatient hospitalization.
- Results in persistent or significant disability or incapacity.
- Is a congenital anomaly or birth defect in the child or fetus of a patient exposed to IP prior to conception or during pregnancy.
- Is an important medical event or reaction.

The reporting period for SAEs begins after informed consent is obtained, and continues until 4 weeks following the last administration of study drug or End of Treatment Visit.

All SAEs, whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form to BioMarin Pharmacovigilance (BPV). ). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the patient's medical record.

For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).

At the last scheduled visit, the Investigator should instruct each subject to report any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study treatment.



The Investigator should notify the study Sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior study treatment. The Sponsor should also be notified if the Investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that participated in this study.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

### 10.3 Pregnancy

Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up Form in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

#### **10.4** Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "... in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours.

|----------|---------|---------|

Examples of situations that may require urgent safety measures include discovery of the following:

- Immediate need to revise the IP administration (ie, modified dose amount or frequency not defined in protocol).
- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.



# 10.5 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the medical monitor any AEs for which the issue of seriousness is unclear or questioned. Contact information for the medical monitor is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:

Fax:

E-mail:



### 11 APPROPRIATENESS OF MEASUREMENTS

# 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

# 11.2 Diet Diary

A 3-day diet diary will be issued to subjects for completion and will be brought to each clinic visit for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6.



#### 12 STUDY PROCEDURES

# 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

# 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- Chest X-ray
- 12-lead ECG
- Clinical laboratory tests (including hematology, chemistry, and urinalysis)
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in PAL-002 or PAL-004, these assessments may be the same as those used for the Week 16 Visit of PAL-002 or the Week 16 visit of PAL-004, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.



If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done daily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

# 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs, including weight
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (postdose)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)
  - For subjects enrolling into this study from Study PAL-004, first dose of rAvPAl-pEG must be given in the clinic setting and a telephone follow-up with the subject must be performed 24 hours later to assess safety issues.



#### 12.3.2 Weekly Visits

Weekly visits do not require an in-clinic visit if conducted by a home healthcare professional. However, dose modifications must be performed in the clinic. Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

The following study activities will be performed at the weekly visits beginning with Week 2:

- Vital signs, including weight
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)
- PK sample
- For subjects participating in the Substudy, refer to Section 12.3.3.
- Blood Phe and plasma tyrosine concentration
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)
  - o For subjects participating in the Substudy, refer to Section 12.3.3.

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.



## 12.3.3 Substudy Visits (Weekly)

The following study activities will be performed on Day 1 of the Substudy (ie, final dose prior to interruption), Day 8, Day 15, Day 22, and Day 29 (ie, restart administration of study drug) for subjects participating in the Substudy:

- Physical examination
- Vital signs, including weight
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (predose; postdose on Day 1; during weekly visit on Day 8, 15, 22; and postdose on Day 29)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies,)
- Blood Phe and plasma tyrosine concentration
  - When dosing is stopped, sampling for blood Phe assessment only will be performed prior to the final dose and then postdose at 8 hours, 12 hours, 16 hours, 24 hours, 48, hours, 72 hours, 96 hours, 144 hours, 168 hours, and 216 hours.
  - When dosing is re-started, sampling for blood Phe assessment only will be performed predose and then postdose at 24 hours, 48 hours, 72 hours, 120 hours, and 168 hours.
- PK sample
- For subjects participating in the Substudy, additional PK sampling will be performed upon the final dose prior to the planned dosing interruption and upon re-introduction of rAvPAL-PEG. Refer to Section 9.7.3
- Administer study drug (Day 29 only)



o For subjects participating in the Substudy, administration of rAvPAL-PEG will not be performed for approximately 4 consecutive weeks regardless of their dosing regimen (dose level and frequency). After approximately 4 weeks of no dosing, rAvPAL-PEG administration will be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of re-administration must be given in the clinic setting, and a telephone follow-up with the subject must be performed 24 hours later to assess safety issues.

# 12.3.4 Monthly Visits (Week 4, 8, 12, etc)

Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Monthly visits consist of all weekly activities and include additional activities and must be performed in the clinic. The following study activities will be performed at the monthly visits beginning with Week 4:

- Vital signs, including weight
- Clinical laboratory tests
- Chest x-ray (Month 12 visit only)
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)
- PK sample
- For subjects participating in the Substudy, refer to Section 12.3.3.
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)



- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)
  - o For subjects participating in the Substudy, refer to Section 12.3.3.

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

# 12.3.5 Quarterly Visits (Week 12, 24, 36, etc)

Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Quarterly visits consist of all weekly and monthly activities and include additional activities. The following study activities will be performed at the quarterly visits beginning with Week 12:

- Physical examination
- Vital signs, including weight
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)
- PK sample
  - o For subjects participating in the Substudy, refer to Section 12.3.3.
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)



For subjects participating in the Substudy, refer to Section 12.3.3.

In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home.

## **12.3.6 Interim Dosing Visit**

Subjects who increase their dose frequency during the study from 1x/week to 2x/week or daily will have additional assessments performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased. If the Interim Dosing Visit coincides with a weekly, monthly, or quarterly scheduled visit, the scheduled visit assessments should also be performed. The following study activities will be performed for the Interim Dosing Visit:

- Vital signs, including weight
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Blood Phe measurement by fingerstick
  - o This may be done by the subject at home.

## 12.3.7 Unscheduled Hypersensitivity Reaction Visit

Subjects who have a systemic reaction, including a generalized skin reaction, or a large local skin reaction that is not contiguous to the injection site after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 48 hours) the reaction.

- Injection-site inspection
- Clinical laboratory tests
- Sedimentation rate
- CRP, CH50, C1, C3, and C4
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies)
- Serum tryptase level
- Perform immediately after reaction if possible.
- Skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction)



- PK sample
- Assessment of AEs
- Concomitant medications

Following completion of the Unscheduled Hypersensitivity Reaction Visit assessments, the subject may resume treatment with study drug per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. Subjects who have had an IgE-mediated reaction must be discontinued from further study drug administration. Subjects who do not have an IgE-mediated reaction may resume study drug administration under close monitoring; subjects must be premedicated orally with acetaminophen and/or antihistamines 1 hour prior to study drug dosing for the remainder of the study (refer to Section 9.1.1.3.3).

### 12.4 Early Termination Visit

The Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug. Subjects who terminate from study treatment early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications



- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)

## 12.5 Final Follow-up Visit

The final follow-up (F/U) Visit will occur 1 week after the final dose of study drug.

The following study activities will be performed at the F/U Visit:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Final Follow-up Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)



# 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

# 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

### 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseine, of vital signs, ECG results, and X-ray results will also be provided.

### 14.3 Pharmacokinetic Analysis

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $C_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F). Should data become available from PAL-002 or PAL-004 that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.



## 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 60-600 µmol/L will be summarized by each scheduled time point.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis. Information regarding this exploratory analysis will be provided in the Statistical Analysis Plan.

For subjects who completed the Substudy, the effect of stopping and re-starting rAvPAL-PEG dosing on safety, blood Phe level, and immune response will be explored. Information regarding the analysis will be provided in the Statistical Analysis Plan.

### 14.5 Determination of Sample Size

Subjects who participated in PAL-002 or PAL-004 may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

### 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.

### 14.7 Interim Analyses

Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

# 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these



circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.



#### 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study. Meetings of the DMC can be convened at any time at the discretion of the DMC Chair or the Study Medical Officer. The Chair will be notified by the Study Medical Officer of all SAEs and will receive summaries of other safety data as available. The DMC will review the study data as soon as it is available during the study, on a schedule defined in the DMC Charter, and offer advice on whether or not to proceed, modify or terminate study enrollment on the basis of toxicity. Details regarding the DMC membership and safety data to be reviewed by members will be provided in a charter.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.3.



# 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment. If the subject has followed the Investigator's instructions, BioMarin will pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures, if these costs are not covered by health insurance or another third party that usually pays these costs. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.



#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent. If an Investigator or institution refuses to allow access to subject records because of confidentiality, arrangements must be made to allow an "interview" style of data verification.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the

|-------------------------------|----------|
|-------------------------------|----------|

clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.



### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (eg, subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.



### 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.



#### 21 REFERENCES

Armstrong, JK, Hempel, G, Koling, S, Chan, LS et. al. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007.

Chen, AM, Scott, MD. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001.

Davis, S, Abuchowski, A, Park, YK, Davis, FF. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981.

Fisch, RO. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000.

Gamez, A, Wang, L, Sarkissian, CN, Wendt, D et. al. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007.

Ganson, NJ, Kelly, SJ, Scarlett, E, Sundy, JS et. al. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006.

Guttler, F, Azen, C, Guldberg, P, Romstad, A et. al. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003.

Harris, JM, Chess, RB. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003.

Huttenlocher, PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000.

Kaufman, S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989.

Koch, R, Hanley, W, Levy, H, Matalon, K et. al. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003.

Lapis. Long-term Correction of PKU in the Pahenu2 Mouse by Mutant and Chemically Modified Forms of Phenylalanine Ammonium Lyase. ASHG 57th Annual Meeting The American Society of Human Genetics)2007.



Lee, PJ, Lilburn, M, Baudin, J. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003.

Levy, HL. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003.

Matalon, R, Surendran, S, Matalon, KM, Tyring, S et. al. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003.

Richter, AW, Akerblom, E. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983.

Richter, AW, Akerblom, E. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984.

Rouse, B, Azen, C. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004.

Scott, MD, Murad, KL, Koumpouras, F, Talbot, M et. al. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997.

Scriver, CR, Kaufman. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-1724.

Walter, JH, White, FJ, Hall, SK, MacDonald, A et. al. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002.

Webster, R, Didier, E, Harris, P, Siegel, N et. al. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007.



#### 22 INVESTIGATOR RESPONSIBILITIES

# 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.

| BIOMARIN° PAL-003 Page 111 |
|----------------------------|
|----------------------------|

#### 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

**Protocol Number: PAL-003** 

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

| Investigator | Signature | Date |
|---------------|-----------|------|
| Printed name: | | |

### Accepted for the Sponsor:

On behalf of BioMarin, I confirm that BioMarin, as a sponsor will comply with all obligations as detailed in all applicable regulations and guidelines. I will ensure that the PI is informed of all relevant information that becomes available during the conduct of this study.

| | , | May 4, 2011 |
|-----------------|---|-------------|
| Medical Monitor | | Date |
| Printed name: | | |




# 24 PROTOCOL AMENDMENT TEXT REVISIONS

The following table summarizes the revisions made to the protocol and relates the changes to the appropriate rationale. Text that has been added or inserted is indicated by underlined font, and deleted text is indicated by strikethrough font.

| Section No./Title | | |
|---|---|---|
| Section 2/Synopsis (Study Sites) | Approximately 208 centers in the United States | 4 |
| Section 2/Synopsis (Study Rationale) | The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. Phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the dose-finding studiesy (Study PAL-002 and Study PAL-004). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects. Because rAvPAL-PEG is being assessed as a long-term chronic treatment for patients with PKU, there is a need to understand the effect of a temporary dosing interruption on the safety, efficacy (blood Phe), PK, and immune response. Therefore, a Substudy has been added to this study to assess the effects of stopping and re-starting rAvPAL-PEG treatment in subjects who are on a variety of rAvPAL-PEG dosing regimens (dose level and frequency). Up to 10 subjects who are on a variety of dosing regimens (dose level and frequency) in this study are eligible for participation in the Substudy and will stop dosing for a period of approximately 4 weeks. During this dosing interruption, subjects will be assessed for safety, efficacy, PK, and immune response and will continue to perform the scheduled study assessments. Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, | 1, 5 |




| Section No./Title | | |
|---|---|---|
| | an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary. | |
| Section 2/Synopsis<br>(Objectives) | <ul> <li>The secondary objectives of the study are: <ul> <li>To evaluate the immune antibody response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.</li> <li>To evaluate steady state PK of rAvPAL PEG in subjects with PKU.</li> </ul> </li> <li>The exploratory objective of the study is as follows: <ul> <li>To assess the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.</li> </ul> </li> <li>The Substudy objectives are as follows: <ul> <li>To assess the safety and tolerability of stopping and re-starting rAvPAL-PEG dosing in a subset of subjects with PKU.</li> </ul> </li> <li>To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on blood Phe concentration in a subset of subjects with PKU.</li> <li>To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on immune response in a subset of subjects with PKU.</li> <li>To assess the effect of multiple doses of rAvPAL-PEG on the PK profile, in particular clearance of drug, when drug is stopped in a subset of subjects with PKU who have been previously exposed to rAvPAL-PEG.</li> </ul> | 1, 5, 14 |
| Section 2/Synopsis (Stud<br>Design and Plan) | This is a long-term extension of athePhase 2, open-label, dose-finding studies,y (Study PAL-002 and PAL-004, in 35–50 approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 51.0 mg/kg/weekper injection), provided no dose-limiting toxicity iwas observed in | 1-4, 6, 27 |

| BIO | M | A | R | N | 8 |
|-----|---|---|---|---|---|
|-----|---|---|---|---|---|


| Section No./Title | |
|---|---|
| | PAL-002 or PAL-004. |
| | Only subjects who completed the protocol-defined study drug regimen participation in PAL-002 or PAL-004 will be enrolled into this study. Subjects who enroll from PAL-002 will either continue the dose regimen that was administered upon completion of PAL-002 or start dosing at a higher dose per the dose increase instructions. Subjects who enroll from PAL-002 may start this study at a higher dose level provided there was no interruption in dosing since completion of PAL-002 and enrollment into this study. Subjects who enroll from PAL-004 will re-start rAvPAL-PEG dosing in this study at the same dose level and frequency as was administered upon completion of PAL-004. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing in this study. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Diet will-should not be altered during the course of this study, except as necessary for safety as determined by blood Phe concentrations. If a subject's blood Phe concentration is < 120 µmol/L, the subject's diet may be adjusted to increase the amount of dietary Phe |
| | intake to maintain target blood Phe concentrations of 120 600 µmol/L. Changes to diet will |
| | be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigaor in consultation with the Sponsor's Medical Officer.To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff. |
| | Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration. |
| | Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 43. |
| | At least one interim analysis may be performed by the sponsor during the study. In addition |

| B <sub>2</sub> OI | MA | RI | N° |
|-------------------|----|----|----|
|-------------------|----|----|----|


| Section No./Title | |
|---|---|
| | to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor. |
| | PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 and PAL-004 subjects' rAvPAL-PEG dosing will continue in PAL-003 without interruption of dosing. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 6120-600 µmol/L. Doses will be evaluated on an individual basis. |
| | Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (6120-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer but not to exceed 3x/week (fingerstick tests may be performed more frequently). |
| | A subject will continue in PAL-003 until one of the following occurs: |
| | The subject withdraws consent and discontinues from the study. |
| | 2. The subject is discontinued from the study at the discretion of the Investigator. |
| | 3. The subject has completed the study through the Month 2460 visit. |
| | 4. The study is terminated. |
| | Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety. |
| | PAL-003 Substudy |
| | A subset of up to 10 subjects who are already enrolled and who have consented to |

| BIO | MA | R | IN |
|-----|----|---|----|
|-----|----|---|----|


| Section No./Title | | |
|---|---|---|
| | participate in this study will be asked to participate in a Substudy to assess the effect that stopping and re-starting treatment with rAvPAL-PEG has on safety, efficacy, PK, and immune response. Subjects will be eligible for participation in the Substudy provided they also meet all of the PAL-003 eligibility criteria, have been on a stable dosing regimen for approximately 4 weeks during this study, have not had any serious adverse events reported during PAL-003, and were not enrolled in Study PAL-004. Subjects participating in the Substudy will have rAvPAL-PEG administration halted for approximately 4 weeks regardless of their dosing regimen (dose level and frequency). rAvPAL-PEG will not be administered during the dose interruption; however, subjects will continue to perform assessments for safety, blood Phe concentration, PK, and immune response. Subjects enrolled into the Substudy will also have additional PK sampling performed prior to the dosing interruption and during the dosing interruption. To allow for PK sampling once dosing is stopped, subjects may be admitted to a research facility within 8 hours of stopping dosing where they will reside for at least 24 hours. After the dosing interruption, rAvPAL-PEG administration will be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. Upon re-starting rAvPAL-PEG, the first dose must be administered in the clinic and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Additional PK sampling will also be performed for the first week after the dosing interruption. | |
| Section 2/Synopsis (Dose Modifications) | Dose Modifications: After any modifications (increases or decreases) to dose level or frequency, subjects should remain in the clinic for observation for at least 2 hours following the injection of study drug. The Investigator should remain at the site to assess the subject for safety. | 2, 3, 21, 22 |
| | Dose Increase Methodology: Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations. Blood Phe levels will be measured 3 days after each dose increase (fingerstick is | |

| BIO | MA | AR | IN° |
|-----|----|----|-----|
|-----|----|----|-----|


| Section No./Title | |
|---|---|
| | acceptable); more frequent or daily blood Phe measurements may be performed. |
| | For subjects from PAL-002 only Depending upon the response to rAvPAL PEG in PAL 002, an individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows. |
| | • The dose may be increased by increments of no more than 10-fold higher than the subject's current dose. |
| | • When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, and 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg) that were defined in the previous study (PAL 002).or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 μmol/L) and drug concentrations, as well as any adverse events (any hypersensitivity reaction) for an individual subject. |
| | • The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 52.0 mg/kg, including subjects who receive more than 1 dose/week. Subjects who increase their dose frequency will have additional assessments performed (Interim Dosing Visit). |
| | • When a dose is increased (either by increasing the dose level or by increasing the frequency of dosing), the subject must remain in the clinie be observed for a minimum of 30-60 minutes 2 hours following the first modified dose administration, and an Investigator will remain on site during this time. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount. |
| | • Only 1 dose ( <u>level or frequency</u> ) adjustment is allowed every 2 weeks. |
| | • Blood Phe levels will be measured <u>daily for</u> 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements |



| Section No./Title | | |
|---|---|---|
| | may be performed. | |
| | Dose Decrease Methodology | |
| | A subject's diet should be assessed prior to any dose decreases. Changes to diet should only be made if a subject's blood Phe concentrations < 120 μmol/L. If a subject's blood Phe level is < 120 μmol/L, the subject's dietary Phe intake should be increased to achieve a stable blood Phe concentration of 120 600 μmol/L. If the subject's blood Phe level is < 120 μmol/L despite a high Phe diet, the rAvPAL PEG dose will then be decreased. The subject will be asked about any changes to diet prior to any dose adjustments, and any changes to diet should be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. | |
| | All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 μmol/L > 30% change from baseline) and drug concentrations, as well as any adverse eventstoxicity (any hypersensitivity reaction). Dose decreases may occur for safety (ie, blood Phe concentration < 120 μmol/L) or other toxicity any adverse event that may be improved with a lower, more frequent dose). | |
| | A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced. | |
| Section 2/Synopsis (Stopping Safety Assessment Criteria) | Safety AssessmentStopping Criteria: If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same | 8 |




| Section No./Title | | |
|---|---|---|
| | dose level, or restart dosing at a lower dose level. | |
| | Stopping Criteria: | |
| | In addition, if 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will be evaluated and halted and no subjects will be treated at a higher dose level until a safety assessment will be is completed. In addition, the Food and Drug Administration (FDA) will-may-be notified of this occurrence if appropriate. | |
| Section 2/Synopsis | 35 50 Approximately 100 subjects. | 4 |
| (Number of Subjects | | |
| Planned) | | |
| Section 2/Synopsis | Individuals eligible to participate in this study must meet all of the following criteria: | 4, 11 |
| (Diagnosis and All Criteria for Inclusion and | <ol> <li>Must have completed participation and all protocol-defined study drug in PAL-<br/>002 or PAL-004.</li> </ol> | |
| Exclusion) | Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study: | |
| | <ol> <li>Use of any investigational product (with the exception of rAvPAL-PEG) or<br/>investigational medical device within 30 days prior to Screening, or<br/>requirement for any investigational agent prior to completion of all scheduled<br/>study assessments.</li> </ol> | |
| | 2. Use of any medication <u>other than rAvPAL-PEG</u> that is intended to treat PKU within 14 days prior to the administration of study drug. | |
| | 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation. | |
| | 4. A prior reaction that included systemic symptoms (eg, generalized hives, | |

| BIO | M | A | R | IN° |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | | |
|---|---|---|
| | respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study. 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL-002 or PAL-004. | |
| Section 2/Synopsis (Investigational Product, Dose, Route, and Regimen) | rAvPAL-PEG doses will be administered SC provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1 mL of the drug product. Upon enrollment into this study, subjects from PAL-002 will be dosed with the same or higher dose than the dose that was administered upon completion of PAL-002. Subjects enrolling from PAL-004, will be administered the same dose that was administered upon completion of PAL-004. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on on available information regarding a subject's blood Phe level (60-600 μmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 6120-600 μmol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. | 1, 3, 4, 27 |
| Section 2/Synopsis | Up to 60 months. Extension of multiple dosing will continue until one of the following | 17 |
| (Duration of Treatment) | occurs: | |




| Section No./Title | | |
|---|---|---|
| | <ol> <li>The subject withdraws consent and discontinues from the study.</li> <li>The subject is discontinued from the study at the discretion of the Investigator.</li> <li>The subject has completed the study through the Month 24 visit.</li> <li>The study is terminated.</li> </ol> | |
| Section 2/Synopsis<br>(Criteria for Evaluation) | Immunogenicity: The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies) | 22, 27 |
| | Safety: Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant | |
| | Pharmacokinetic: Plasma concentrations of rAvPAL-PEG will be measured when steady state levels of Phe | |
| 2. The subject is discontinued from the study at the discretion of the Investigator. 3. The subject has completed the study through the Month 24 visit. 4. The study is terminated. 22, 2 Immunogenicity: The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgG, anti-PEG IgG, and anti-rAvPAL-PEG neutralizing antibodies) will be assessed. Safety: Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs, ECG results, X-ray results, and or laboratory test results. Pharmacokinetic: Plasma concentrations of rAvPAL-PEG will be measured when steady state levels of Phe are attained for subjects participating in the Substudy. | 1, 3, 4, 5, 27 | |
| • • | Subjects who participated in PAL-002 or PAL-004 may be enrolled into this study. | -, -, -, -, -, |
| | Safety Analysis: | |




| Section No./Title | |
|---|---|
| | subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Safety will be evaluated on the incidence of AEs, including serious AEs (SAEs), and clinically significant changes in vital signs and laboratory test results. Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, ECG results, and X-ray results will also be provided. |
| | Efficacy Analysis: |
| | Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis. |
| | Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 12060-600 µmol/L will be summarized by each scheduled time point. |
| | Exploratory Analysis: |
| | For subjects who have received any study drug in this study with any post-treatment blood Phe concentration measurements and diet diary information, the relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will be explored. |
| | Substudy Analysis: |
| | For subjects who completed the Substudy, the effect of stopping and re-starting rAvPAL-PEG dosing on safety, blood Phe level, and immune response will be explored. |




| Section No./Title | | |
|---|---|---|
| | Pharmacokinetic Analysis: | |
| | Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis. | |
| | Steady state PK (predose samples) of rAvPAL PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (120-600 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Should data become available from PAL 002 that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed rbut not to exceed 3x/week. | |
| | Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration $(T_{max})$ , maximum plasma concentration $(C_{max})$ , half life $(t_{1/2})$ , and clearane $(CL/F)$ . | |
| Tables 2.1/Schedule of | Table 2.1.1, Schedule of Events, has been revised to reflect change made to the study. | 13, 16, 18, |
| Events | Table 2.1.2, Schedule of Events-Substudy, has been added. | 19, 22, 23, |
| | Tables 2.1.23 and 2.1.34, Interim Dosing Visit Schdules, have been revised to remove the PK sampling. | 24, 26 |
| Section 4/List of | C <sub>3</sub> complement 3 | 27 |
| Abbreviations and Definitions of Terms | C <sub>4</sub> complement 4 | |
| 2 | rAvPAL-PEG rAv recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG | |
| Section 6/Investigators and | Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase | 27 |
| Administrative Structure | polyethylene glycol (rAvPAL and rAvPAL-PEG) IgE antibody analysis will be performed | |
| | by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory | |
| | tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a | |

| BIO | MA | RI | N° |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| | central laboratory, with the exception of erythrocyte sedimentation rate (ESR), urinalysis, | |
| | and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A | |
| | central laboratory will also be used to perform analysis of blood phenylalanine (Phe) | |
| | concentrations. Pharmacokinetic (PK) analysis will be performed by BioMarin. | |
| Section 7.1/Nonclinical | The nonclinical program for rAvPAL-PEG has characterized the pharmacology, | 1, 25 |
| Studies | pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC | |
| | route of administration. Pharmacology was assessed in the BTBR <i>Pah</i> <sup>enu2</sup> (ENU2) mouse | |
| | model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU | |
| | patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to | |
| | 2000 μM) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to | |
| | male ENU2 mice, plasma Phe concentrations decreased from approximately 2000 μM to | |
| | < 200 μM after 2 dose administrations. An attenuated reduction of blood Phe was seen | |
| | between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, | |
| | pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe | |
| | < 200 μM over the entire week, which continued for a total of 15 weeks. | |
| | In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered | |
| | 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a | |
| | 2-4 week dose interruption and an 11-week dose interruption. Following both dose | |
| | interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. | |
| | No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily | |
| | stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A | |
| | similar interim attenuated response was observed with the longer dose interruption of | |
| | approximately 11 weeks. In both of these assessments, no safety issues were noted upon | |
| | re-starting dosing with rAvPAL-PEG (Lapis et al., Long-term correction of PKU in the | |

| BIO | M | A | R | IN° |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | |
|---|---|
| Section 140./ Title | |
| | Pahenu2 mouse by mutant and chemically modified forms of Phenylalanine Ammonium |
| | Lyase. The American Society of Human Genetics, 57th Annual Meeting, 2007). |
| | Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No |
| | respiratory or central nervous system (CNS) effects were seen with SC administration of |
| | rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram |
| | (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV |
| | effects of rAvPAL-PEG administered subcutaneously. |
| | Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats |
| | and cynomolgus monkeys. The elimination half-life (t <sub>1/2</sub> ) values of rAvPAL-PEG |
| | administered to normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and |
| | 44 hours, respectively, and exhibited modest area under the plasma concentration-time |
| | curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, |
| | the t <sub>1/2</sub> was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 |
| | mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey |
| | appear to have similar characteristics. The following findings were noted: (1) a |
| | 1-compartment model with first-order absorption appears to describe the plasma profiles of |
| | rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long |
| | absorption period after SC administration to maximum observed plasma concentration |
| | ( $C_{max}$ ), along with a long $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not |
| | appear to be a gender difference, and (5) the AUC and the $C_{max}$ are roughly linearly |
| | proportional. |
| | Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal |
| | rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and |
| | Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the |
| | Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a |


## Section No./Title 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given ≥ 3 mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey. The murine model of phenylketonuria (PKU) BTBRPah (ENU2), a mouse line that is deficient in phenylalanine hydroxylase (PAH) activity (Shedlovsky, 1993, Genetics), was used for in vivo screening and pharmacodynamic studies. This mouse model exhibits characteristics similar to those seen in PKU patients, including hyperphenylalaninemia (baseline plasma phenylalanine [Phe] concentrations of 1000 to 2000 μM) and hypopigmentation. Weekly subcutaneous (SC) administration of 80 mg/kg of rAvPAL PEG (approximately 4 IU/mouse) for greater than 2 to 3 months lowered and stabilized plasma Phe concentration from approximately 2000 µM to less than 200 µM. A similar profile of Phe reduction was also seen in ENU2 mice administered wild type AvPAL PEG (4 IU/mouse) over 8 weeks. In all these studies, regardless of the molecule, an attenuated Phe lowering response was usually seen between Weeks 2 and 7. However, plasma Phe concentrations became stable at concentrations below 200 µM from Week 7 onward. In addition to the reduction of plasma Phe, a dose related darkening in coat color occurred,


| Section No./Title | | |
|---|---|---|
| | indicating the biosynthesis of melanin, which was previously inhibited when plasma Phe | _ |
| | could not be metabolized and plasma Phe concentrations were high. When administration of | |
| | AvPAL PEG was stopped for 2 to 7 weeks and then reinitiated with weekly | |
| | administrations, no attenuated response was observed and Phe concentrations remained low | |
| | and stable until the next administration. | |
| | The safety of rAvPAL PEG was evaluated in safety pharmacology studies (respiratory, | |
| | central nervous system [CNS] and cardiovascular [CV]) and toxicity with toxicokinetic | |
| | studies (single and 28 day repeated dose) in rats and cynomolgus monkeys. Overall, in the | |
| | nonclinical studies, no anaphylactoid like reactions or injection site reactions were noted. | |
| | No specific polyethylene glycol (PEG) related histological findings were observed during | |
| | the 28 day repeated dose studies. | |
| | Findings in cynomolgus monkeys dosed with a single administration of | |
| | 60 mg/kg rAvPAL PEG included reduced food consumption, dehydration, body weight | |
| | loss, hypoactivity, hypothermia, decreased plasma Phe concentration, decreased protein | |
| | synthesis, and gastrointestinal (GI) lesions. Plasma Phe concentrations were also reduced to | |
| | below the level of detection in the 4 and 12 mg/kg dose groups, but without similar | |
| | toxicological consequences, implying that the physiological regulation of Phe levels may be | |
| | an important factor for influencing morbidity. | |
| | The main finding in the 28 day study was the possible drug related observation of minimal | |
| | to slight degeneration of blood vessels of predominantly medium sized muscular arteries | |
| | with a non-dose dependent involvement of different organs observed in 1 male in the | |
| | 0.1 mg/kg and 1 male and 1 female in the 1.0 mg/kg rAvPAL PEG dose groups. No | |
| | degeneration of the arteries was observed in either the control or animals administered 0.01 | |
| | mg/kg rAvPAL PEG. | |
| | The half life of rAvPAL PEG administered to normal rats at SC doses of 10, 25, and | |


## Section No./Title 250 mg/kg, was 47, 33, and 44 hours, respectively, and exhibited modest area under the plasma concentration time curve (AUC) dose linearity. In the cynomolgus monkey after SC administration of rAvPAL PEG, the half life was 65 hours at 4 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1 compartment model with first order absorption appears to describe the plasma profiles of rAvPAL PEG after single dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum plasma concentration, along with a long half life, (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) AUC and the maximum plasma concentration (C<sub>max</sub>) are roughly linearly proportional. Chronic repeat dose toxicity and toxicokinetic studies were conducted in the rat (17/26 weeks) and monkey (39 weeks). In the 26 week study of rats, weight loss was observed in the rats given 25 mg/kg/dose of rAvPAL PEG, SC; corresponding decreased food consumption was observed in the males. The main histological finding was focal to multifocal areas of vacuolar degeneration of renal tubule cells in the kidney of 3 males given 25 mg/kg and 3 females given ≥ 8 mg/kg rAvPAL PEG. This renal tubule finding persisted in the kidney of both sexes given ≥ 8 mg/kg/dose at the end of the 12 week recovery phase without evidence of reversibility. Increased vacuolation was observed in histiocytic cells of the liver, spleen, mesenteric lymph node, mandibular lymph node, and adrenal cortex of males given 25 mg/kg/dose and females given ≥ 8 mg/kg/dose; vacuolation of histiocytic cells in the testes were also observed in males given 25 mg/kg/dose. Both renal tubule vacuolation and histiocytic cell vacuoles have been associated with PEG related catabolism and administration of other PEGylated proteins. In the 39 week, chronic repeat dose toxicity and toxicokinetic study in monkeys, dose

| BIO | M | A | R | IN. |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | | |
|---|---|---|
| | levels of 7.0 and 5.0 mg/kg/dose rAvPAL PEG were not tolerated in female monkeys and | |
| | resulted in body weight loss, decreased food consumption, and hypoactivity. The only | |
| | adverse microscopic finding was arterial inflammation of small and mid sized arteries in | |
| | multiple organs and/or tissues in most animals that were given ≥ 3 mg/kg/dose rAvPAL | |
| | PEG SC twice weekly at the end of the dosing phase. The inter individual organ | |
| | involvement was highly variable; some animals had findings in one organ and others had | |
| | multiple organs with arterial inflammation. Additionally, not all arteries had signs of | |
| | inflammation and arterial inflammation was resolved by the end of the 13 week recovery | |
| | period. A full analysis of these findings including the involvement of the anti-drug | |
| | antibodies, antibody isotypes, PEG distribution, and rAvPAL PEG is ongoing. The no | |
| | observable adverse effect level (NOAEL) for the 17 week and 39 week studies, in rat and | |
| | monkey, respectively, is 1 mg/kg/dose. The NOAEL from these studies represents greater | |
| | than a 100 fold safety factor over the starting dose in PAL 002. | |
| Section 7.2/Previous | This study is an extension of the second human clinical study with rAvPAL PEG | 20 |
| Clinical Studies | (Study PAL 002). Study PAL 001, the first in human clinical study of rAvPAL PEG, was | |
| | designed as a Phase 1, open label, single dose, dose escalation study in 25 subjects, 16 to | |
| | 50 years old, with PKU. The doses for this study are based on data from nonclinical studies | |
| | and PAL 001 and are 0.001 through 1.0 mg/kg per injection (not to exceed 2.0 mg/kg/week, | |
| | provided no dose limiting toxicity was observed in Study PAL 002. | |
| | The rAvPAL-PEG clinical development program has been designed to demonstrate the | |
| | safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU patients | |
| | who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. | |
| | This study is an extension of the ongoing human clinical studies with rAvPAL-PEG | |
| | (Study PAL-002 and Study PAL-004) based on data from the completed clinical study, | |

| B.C | MA | RI | N |
|-----|----|----|---|
|-----|----|----|---|


| Section No./Title | | |
|---|---|---|
| | PAL-001, and clinical experience to date (JAN2011) from this ongoing study and the other ongoing Phase 2 study, PAL-002, and are 0.001 through 5.0 mg/kg/week. | |
| Section 7.2.1/Phase 1<br>Study: PAL-001 | The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations. The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 μmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG. Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows: • rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg. • For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, | 20 |

| BIO | MA | \R | IN. |
|-----|----|----|-----|
|-----|----|----|-----|


| Section No./Title | | |
|---|---|---|
| | <ul> <li>0.01, and 0.03 mg/kg.</li> <li>For subjects who were administered rAvPAL-PEG at the 3 higher dose levels (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration levels, the calculated PK parameters were a mean T<sub>max</sub> of 89-106 hours, a t<sub>1/2</sub> of 46-120 hours, and an AUC<sub>0-t</sub>, and C<sub>max</sub> that were proportional with dose. Drug exposure was slightly increased with increased dose.</li> </ul> | |
| Section 7.2.2/Phase 2<br>Studies: PAL-002 and<br>PAL-004 | Currently, rAvPAL-PEG is being investigated in two Phase 2 clinical trials (PAL-002 and PAL-004). To date (JAN2011), a total of 33 subjects have been administered rAvPAL-PEG in Study PAL-002 and initiation and recruitment of clinical sites is underway for Study PAL-004. In PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU), approximately 55 subjects will be enrolled and will be administered multiple doses of rAvPAL-PEG up to 5.0 mg/kg/week. PAL-002 is a 2-part study. In Part 1, subjects will be assigned to 1 of 4 rAvPAL-PEG dose cohorts (0.001, 0.003, 0.01, 0.1 mg/kg, or 1.0 mg/kg). rAvPAL-PEG will be administered at a fixed weekly dose of 0.001 mg/kg (Cohort 1), 0.003 mg/kg (Cohort 2), 0.01 mg/kg (Cohort 3), 1.0 mg/kg (Cohort 4), or 0.1 mg/kg (Part 1 Substudy) for 8 weeks. In Part 2, all subjects who complete Part 1 will be administered an adjustable dose of rAvPAL-PEG for up to an additional 8 weeks. The dose administered in Part 2 may be adjusted by dose level and/or dose frequency to reach a target blood Phe concentration of 60-600 μmol/L. Study PAL-003 (Long-Term Extension of a Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU) is an extension study of PAL-002 and PAL-004. Once subjects have completed Study PAL-002 or PAL-004, they have the option to enroll into PAL-003 and to continue to receive doses of rAvPAL-PEG | 20 |

| BIO | MA | RI | N° |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | |
|---|---|
| | for up to an additional 60 months. |
| | Study PAL-002 was initiated in September 2009 and is ongoing. The primary objective of |
| | this study is to evaluate the effect of multiple doses of rAvPAL-PEG on blood Phe |
| | concentrations in subjects with PKU for up to 16 weeks of treatment. The secondary |
| | objectives of the study are (1) to evaluate the safety and tolerability of SC injections of |
| | multiple dose levels of rAvPAL-PEG, (2) to evaluate the antibody response to rAvPAL- |
| | PEG, and (3) to evaluate the PK profile of rAvPAL-PEG in subjects with PKU. The study |
| | protocol was amended (30APR2010) to include a substudy of an additional rAvPAL-PEG |
| | dose level (0.1 mg/kg/week) that reduced blood Phe concentrations to clinically significant |
| | levels in the Phase 1 study, PAL-001. The protocol was amended again (28MAR2011) to |
| | increase the starting dose for Cohort 4 from 0.03 mg/kg/week to 1.0 mg/kg/week. To date |
| | (JAN2011), 33 subjects have been enrolled into the study and all 10 subjects of the |
| | substudy have been dosed with 0.1 mg/kg rAvPAL-PEG. Additional information about the |
| | safety reported to date (JAN2011) is provided in Section 7.4.2. |
| | Study PAL-004 is designed to determine if daily administration of rAvPAL-PEG at daily |
| | dose levels (0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day) is safe and effective in reducing and |
| | maintaining consistent blood Phe concentrations in subjects with PKU. It is hypothesized |
| | that a higher starting dose and frequency will reduce blood Phe concentrations to |
| | near-normal levels in a timely manner and will provide the greatest clinical benefit. |
| | Considering the concentration and volume of drug that is administered subcutaneously, the |
| | only way to increase the rAvPAL-PEG dose is via daily administration. Therefore, in Study |
| | PAL-004, a higher starting dose of 0.4 mg/kg will be administered 5 days a week (referred |
| | to as daily), a dosing regimen that has been observed to be tolerated and to reduce blood |
| | Phe concentrations to clinically meaningful levels in previously exposed subjects in this |
| | study. Following completion of Study PAL-004, subjects have the option to enroll into this |

| BIO | MA | RI | N° |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| | study and to continue to receive doses of rAvPAL-PEG for up to an additional 60 months. | |
| | In this study, subjects in PAL-002 and PAL-004 will continue to be administered the same | |
| | rAvPAL-PEG that was administered in PAL-002 or PAL-004. If the safety, PK, and blood | |
| | Phe concentration results from either PAL-002 or PAL-004 indicate that the appropriate | |
| | level of PEGylation and dosing regimen differs from that administered in PAL-002 or | |
| | PAL-004, the PEGylation and/or dosing regimen administered in this study may change. | |
| Section 7.3/Study | Because rAvPAL-PEG is being assessed as a long-term chronic treatment for patients with | 1, 5 |
| Rationale | PKU, there is a need to understand the effect of a temporary dosing interruption on the | |
| | safety, efficacy (blood Phe), PK, and immune response. To date (JAN2011), there is limited | |
| | information on the effects of a rAvPAL-PEG dose interruption in subjects with PKU. | |
| | Therefore, a Substudy has been added to this study to assess the effects of stopping and re- | |
| | starting rAvPAL-PEG treatment in subjects who are on a variety of rAvPAL-PEG dosing | |
| | regimens (dose level and frequency). Up to 10 subjects who are on a variety of dosing | |
| | regimens (dose level and frequency) in this study are eligible for participation in the | |
| | Substudy and will stop dosing for a period of approximately 4 weeks. During this dosing | |
| | interruption, subjects will be assessed for safety, efficacy, PK, and immune response and | |
| | will continue to perform the scheduled study assessments. There is no information | |
| | regarding the pharmacokinetic (PK) profile of rAvPAL-PEG when blood Phe levels are at | |
| | 60-600 μmol/L for subjects on a multiple-dose regimen. To address this lack of | |
| | information, additional PK sampling will be performed prior to the dosing interruption. | |
| | Upon restarting rAvPAL-PEG, PK sampling will also be performed to allow for collection | |
| | of drug exposure data (area under the plasma concentration-time curve [AUC] and | |
| | maximum plasma concentration [C <sub>max</sub> ]), absorption rate, and clearance for subjects who | |
| | have been previously exposed to rAvPAL-PEG in this Substudy. This information will | |




| Section No./Title | | |
|---|---|---|
| | allow for comparisons to be performed with subjects who were naïve to previous rAvPAL-PEG treatment from the Phase 1 study, PAL-001. Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary. This study is an extension of the dose-finding studiesy (PAL-002 and PAL-004). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of | |
| Section 7.4/Summary of<br>Overall Risks and Benefits | rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects. It is not expected that data from PAL-002 or PAL-004 will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. | 4 |
| Section 7.4.1/Toxicitity Due to Exposure to PEG | Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg | 25 |


| Section No./Title | | |
|---|---|---|
| | rAvPAL-PEG SC. <u>In rats</u> , both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1). | |
| Section 7.4.2/Toxicity Due to an Immunologic Reactions | In Study PAL-001, there were 11 subjects (out of 25 subjects in the study) with skin-related reactions (injection-site bruising, erythema, pain, rash, swelling, and urticaria) that occurred following the single administration of rAvPAL-PEG. For all of these subjects, the reactions were generalized skin reactions or injection-site skin reactions that did not compromise other organs and were not life-threatening. These suspected antibody-mediated responses were nonserious and mild or moderate in severity. These subjects are not considered to be at significant risk for antibody-mediated reactions with injection of rAvPAL-PEG during PAL-002, PAL-004, or this study; however, specific precautions for these subjects will be taken during this study to monitor subject safety (refer to Section 9.1.1). In Study PAL-002, 33 subjects have been dosed to date (JAN2011), including at dose levels of 2.0 mg/kg/week (or 0.4 mg/kg/5 days a week). Most reactions reported in these subjects have been nonserious and mild or moderate in severity. There has been 1 SAE reported to date; the event was reported as not related to treatment with study drug. There have been no reports of anaphylaxis to date (JAN2011). Subjects who have a systemic reaction during this study will undergo a series of assessments to monitor safety, including assessment of IgE antibodies, prior to determining if dosing may resume. Additionally, subjects who have systemic reactions will be premedicated and will be monitored closely for safety (refer to Section 9.1.6 for additional information regarding continued treatment of subjects with systemic reactions during the study). | 9, 11 |

| BIO | MA | AR | IN° |
|-----|----|----|-----|
|-----|----|----|-----|


| Section No./Title | | |
|---|---|---|
| Section 7.4.2.1/Systemic | Two out of 25 subjects who were enrolled in Study PAL-001 and received the | 11 |
| Skin Reactions | protocol-defined single dose of rAvPAL-PEG reported systemic skin reactions (generalized | |
| | skin rash) that were attributed to treatment with study drug. One subject received a single | |
| | dose of 0.001 mg/kg rAvPAL-PEG, and the other subject received a single dose of | |
| | 0.01 mg/kg rAvPAL-PEG. Both of these events were reported as serious and followed | |
| | administration One of these events was reported as serious, and the other was reported as | |
| | nonserious; both events were reported following administration of Depo-Provera injections | |
| | (medroxyprogesterone injection), an injectable contraception. These allergic reactions are | |
| | thought to be related to the PEG molecules that are found in both the study drug, rAvPAL- | |
| | PEG, and Depo-Provera. These reactions are not likely to be experienced concurrent with | |
| | other birth control medications. | |
| | The 2 subjects were administered study drug during PAL-001 and then experienced an | |
| | allergic reaction following an injection of Depo-Provera. The symptoms of the reactions | |
| | were hives on the arms and legs and difficulty breathing. The symptoms for both subjects | |
| | resolved within 1 day following treatment with medication, including the | |
| | . Both subjects were examined by an allergy specialist after | |
| | they completed participation in PAL-001. A skin prick test with Depo-Provera was | |
| | administered as part of this examination. One subject had a mild allergic reaction to the test; | |
| | however, no further reactions or complications were reported following subsequent | |
| | administration of a full dose of Depo-Provera. The Upon study completion, the subject | |
| | continue <u>ds</u> to receive regular doses (every 3 months) of Depo-Provera, and no further | |
| | reactions have been were reported to-date (15OCT2009). The second subject also had a | |
| | positive reaction to Depo-Provera following administration of the skin prick test. When a | |
| | subsequent full dose of Depo-Provera was administered, developed hives, itching, and | |
| | chills. The subject's symptoms resolved within 1 day of taking medication prescribed by an | |


| Section No./Title | | |
|---|---|---|
| Section No./Title | allergist. See Section 7.2.1 for the results from Study PAL-001. The active drug substance in rAvPAL-PEG is a bacterial protein that may elicit immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and others. It is possible that the physio chemical properties of rAvPAL PEG may induce immunologic sensitization to the protein rAvPAL and to PEG. The results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys indicated the formation of anti-rAvPAL antibody titers that did not correspond with observations of injection-site reactions. Quantitation of anti-PEG titers were not assessed in the chronic repeat-dose studies in the rat and monkey. Although results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys did not indicate signs of immune-mediated toxicities, it is possible that the physio-chemical properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG in humans. It is currently unknown whether administration of PEG-containing drugs, such as Depo-Provera, has a sensitizing effect to PEG in rAvPAL-PEG when administered in humans. Because the exact basis for these reported events and their duration is not known, the use of PEG-containing injectable drugs prior to, during, and after this study is prohibited as a precautionary measure (refer to Section 9.3.2 and Section 9.4.8.). | |
| Section | Allergic reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in | 21 |
| 7.4.2.2/Management of Allergic Reactions | intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 230-60 minuteshours post-injection. Longer observations may be required at the discretion of the | |
| | PI. The responsible physician should use all appropriate measures for the treatment of allergic reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the | |

| BIO | M | A | R | IN. |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | | |
|---|---|---|
| | rAvPAL-PEG injection. <u>Subjects who qualify for self administration of study drug will be</u> <u>provided with emergency resuscitation instructions (refer to Section 9.4 and the Subject Self-Administration Training Materials</u> ). | |
| | In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for antibody testing. This additional testing may occur up to 6 months following the final study visit. | |
| | The following measures are recommended for the treatment of allergic symptoms: | |
| | • Clearing Maintain the airway. | |
| Section 7.4.3/Effects of<br>Stopping and Re-Starting<br>rAvPAL-PEG Treatment | The effects of starting, stopping, and re-starting rAvPAL-PEG dosing on safety and blood Phe reductions previously achieved through rAvPAL-PEG dosing are not well defined, and there is limited clinical experience with rAvPAL-PEG. Allergic reactions are a common | 1 |
| | and expected clinical outcome of re-starting biologic drugs, such as rAvPAL-PEG, and may occur when subjects re-start rAvPAL-PEG dosing. However, no information reported from the ongoing clinical studies, including this study, or nonclinical results point to an increased safety risk or decreased efficacy when rAvPAL-PEG dosing is stopped and then re-started | |
| | <ul> <li><u>Nonclinical experience in the the BTBR Pahenu2</u> (ENU2) mouse model indicates that dosing interruptions of 2-4 weeks for mice administered rAvPAL-PEG 80 mg/kg/week had no increased safety risk upon re-starting dosing and there was an immediate return to stable blood Phe reductions (refer to Section 7.1). </li> <li>Antibody results from the ongoing Phase 2 study, PAL-002, and this ongoing study</li> </ul> | |
| | to date (JAN2011) have not indicated an immune response that points to an | |


| Section No./Title | |
|---|---|
| | increased safety risk or decreased efficacy upon re-introduction of drug. There has |
| | not been any immediate immunoglobulin E (IgE)-mediated reactions to rAvPAL- |
| | PEG observed following administration of a rAvPAL-PEG injection. All reactions |
| | to rAvPAL-PEG have been reported approximately 12-24 hours following |
| | administration. To date, 1 out of 33 subjects has tested positive by serology to IgE |
| | antibodies without reporting any clinical symptoms to suggest anaphylaxis or a |
| | severe systemic reaction. Thus, it is not anticipated that reactions to rAvPAL-PEG |
| | are IgE-mediated. |
| | To date (JAN2011), the clinical experience with re-starting rAvPAL-PEG dosing |
| | for subjects from Study PAL-001 who rolled over into Study PAL-002 does not |
| | indicate an increased safety risk or a decreased effect on reducing blood Phe levels |
| | upon re-introduction of drug. |
| | Nine subjects who received a single dose of rAvPAL-PEG and completed |
| | the Phase 1 study, PAL-001, rolled over into the multiple-dose, Phase 2 |
| | study, PAL-002. After a period of several months during which no drug |
| | was administered, these 9 subjects re-started rAvPAL-PEG dosing in Study |
| | PAL-002 at the same starting doses as was administered in Study PAL-001. |
| | There has been no difference to date in the safety profile or efficacy profile |
| | of the subjects from Study PAL-001 who rolled over into Study PAL-002 |
| | (previously exposed to rAvPAL-PEG) when compared with subjects who |
| | were naive to rAvPAL-PEG dosing in Study PAL-002. Although |
| | previously exposed subjects had higher and a faster return of anti-PAL and |
| | anti-PEG IgG titers than those of naïve subjects, these results have not been |
| | associated with a higher safety risk or efficacy riskbased on information to |
| | date. |

| BIO | MA | R | IN. |
|-----|----|---|-----|
|-----|----|---|-----|


| Section No./Title | | |
|---|---|---|
| | o In Study PAL-002, 4 subjects to date have had a protocol-defined (per | |
| | Protocol Amendment # 3 dated 30APR2010), 2-week washout (no dose | |
| | administered) following several weeks of a fixed dose of 0.06 mg/kg/week | <u>ek</u> |
| | or 0.1 mg/kg/week rAvPAL-PEG. Following the 2 weeks where no dose | _ |
| | was administered, all 4 subjects re-started rAvPAL-PEG dosing at a high | er |
| | dose with no safety issues reported to date. Blood Phe levels for these 4 | _ |
| | subjects have not changed upon re-introduction of dosing. | |
| | <ul> <li>Clinical experience with subjects who have had to temporarily halt dosin</li> </ul> | g |
| | due to an adverse event also provides information that stopping and | |
| | re-starting rAvPAL-PEG dosing does not appear to increase the risk to | |
| | subject safety. To date, 10 subjects participating in either PAL-002 or PA | <u>.L-</u> |
| | 003 have had to temporarily stop dosing due to an adverse event. All 10 | |
| | subjects resumed dosing following resolution of the event or per | |
| | determination by the Investigator that subject safety would not be | |
| | jeopardized with re-starting dosing. These 10 subjects resumed dosing at | <u>a</u> |
| | reduced dose level after approximately 1-7 weeks of no dosing. Upon re- | <u>:</u> |
| | starting dosing, none of these 10 subjects have experienced additional | |
| | safety issues. Eight subjects continue to receive dosing with rAvPAL-PE | <u>G</u> |
| | (APR 2011) and have subsequently increased their dose level without | |
| | additional reported adverse events that have resulted in a subsequent dos | ing |
| | interruption. | |
| | In this study, measures will be taken to reduce the risk to subject safety upon re-starting | |
| | rAvPAL-PEG dosing while still allowing for reductions in blood Phe level to clinical | |
| | significance (blood Phe reduction to 60-600 μmol/L). To mitigate the possible safety risk | <u>s</u> |




| Section No./Title | | |
|---|---|---|
| | upon re-starting rAvPAL-PEG dosing, re-introduction of dosing should be performed in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call should be made to subjects 24 hours following re-starting of dosing to monitor subject safety. Subjects will also continue to be assessed per the safety assessment and stopping criteria defined in Section 9.1.3 and Section 9.1.4, and dose decreases will continue to be performed relative to safety as defined in Section 9.1.2.2. To mitigate the possible reduced effect on blood Phe level upon re-starting rAvPAL-PEG, subjects in this study who interrupt dosing whether per the protocol (ie, subjects participating in the Substudy; refer to Section 9.1) or for other reasons (refer to Section 9.4.10) will re-start rAvPAL-PEG dosing at the same dose level. | |
| Section 7.4.3/Effects of | Insufficient Phe intake or excessive rAvPAL PEG exposure may cause blood Phe | 9 |
| Low Blood Phe | concentrations to be too low (eg, < 30 µmol/L). Prolonged low blood Phe concentrations can result in a catabolic state associated with poor growth and altered body functions, including mental and physical alterations, loss of appetite, anemia, rashes, and diarrhea. To ensure safety during this study, subjects will be monitored closely with frequent blood Phe concentration determinations. If a subject's blood Phe concentration is too low, the subject's diet, current dose of study drug, or both may be adjusted. | |
| Section 8/Study Objectives | <ul> <li>The secondary objectives of the study are: <ul> <li>To evaluate the immune antibody response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.</li> <li>To evaluate steady state PK of rAvPAL PEG in subjects with PKU.</li> </ul> </li> <li>The exploratory objective of the study is as follows: <ul> <li>To assess the long-term relationship of diet and change in blood Phe concentration</li> </ul> </li> </ul> | 1, 5, 14 |

| BIO | MA | R | IN° |
|-----|----|---|-----|
|-----|----|---|-----|


| Section No./Title | | |
|---|---|---|
| | <ul> <li>following administration with rAvPAL-PEG in subjects with PKU.</li> <li>The Substudy objectives are as follows: <ul> <li>To assess the safety and tolerability of stopping and re-starting rAvPAL-PEG dosing in a subset of subjects with PKU.</li> <li>To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on blood Phe concentration in a subset of subjects with PKU.</li> </ul> </li> <li>To evaluate the effect of stopping and re-starting rAvPAL-PEG dosing on immune response in a subset of subjects with PKU.</li> <li>To assess the effect of multiple doses of rAvPAL-PEG on the PK profile, in particular clearance of drug, when drug is stopped in a subset of subjects with PKU who have been previously exposed to rAvPAL-PEG.</li> </ul> | |
| Section 9.1/Overall Study Design and Plan | This is a long-term extension of athePhase 2, open-label, dose-finding studies,y (Study PAL-002 and PAL-004, in 35-50 approximately 1000 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 51.0 mg/kg/weekper injection), provided no dose-limiting toxicity iwas observed in PAL-002 or PAL-004. Only subjects who completed the protocol-defined study drug regimen participation in PAL-002 or PAL-004 will be enrolled into this study. Subjects who enroll from PAL-002 will either continue the dose regimen that was administered upon completion of PAL-002 or start dosing at a higher dose per the dose increase instructions. Subjects who enroll from PAL-002 may start this study at a higher dose level provided there was no interruption in dosing since completion of PAL-002 and enrollment into this study. Subjects who enroll from PAL-004 will re-start rAvPAL-PEG dosing in this study at the same dose level and frequency as was administered upon completion of PAL-004. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing in this study. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. | 1-4, 6, 27 |




| Section No./Title | |
|---|---|
| | Diet will-should not be altered during the course of this study, except as necessary for safety as determined by blood Phe concentrations. If a subject's blood Phe concentration is < 120 µmol/L, the subject's diet may be adjusted to increase the amount of dietary Phe intake to maintain target blood Phe concentrations of 120 600 µmol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. For information regarding changes to diet for safety and decreases in dose, refer to Section 9.1.2.2. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigaor in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff. |
| | Subjects may self administer study drug at home if approved by the Sponsor's Medical Officer and if adequate training is provided. Subjects must meet a set of criteria to be considered appropriate for self administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self administration. Additional information is provided in the Subject Self-Administration Training Materials. Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. |
| | Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version <u>43</u> . At least one interim analysis may be performed by the sponsor during the study. In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor. |
| | PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL-002 and PAL-004 subjects' rAvPAL-PEG dosing will continue in PAL-003 without interruption of dosing. In PAL-003, each subject's dose will be adjusted as |




| Section No./Title | |
|---|---|
| | needed to attain or maintain blood Phe concentrations of <u>612</u> 0-600 μmol/L. Doses will be evaluated on an individual basis. |
| | Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 2.1.1, <u>Table 2.1.2</u> , <u>Table 2.1.3</u> , and <u>Table 2.1.4</u> (Schedule of Events). After the subject's blood Phe concentration has been controlled to within a target range (6120-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.but not to exceed 3x/week (fingerstick tests may be performed more frequently). |
| | A subject will continue in PAL-003 until one of the following occurs: |
| | 1. The subject withdraws consent and discontinues from the study. |
| | 2. The subject is discontinued from the study at the discretion of the Investigator. |
| | 3. The subject has completed the study through the Month 2460 visit. |
| | 4. The study is terminated. |
| | Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety. |
| | A subset of up to 10 subjects who are already enrolled and who have consented to participate in this study will be asked to participate in a Substudy to assess the effect that stopping and re-starting treatment with rAvPAL-PEG has on safety, efficacy, PK, and |
| | immune response. Subjects will be eligible for participation in the Substudy provided they |




| Section No./Title | | |
|---|---|---|
| | also meet all of the PAL-003 eligibility criteria, have been on a stable dosing regimen for | |
| | approximately 4 weeks during this study, have not had any serious adverse events reported | |
| | during PAL-003, and were not enrolled in Study PAL-004. Subjects participating in the | |
| | Substudy will have rAvPAL-PEG administration halted for approximately 4 weeks | |
| | regardless of their dosing regimen (dose level and frequency). rAvPAL-PEG will not be | |
| | administered during the dose interruption; however, subjects will continue to perform | |
| | assessments for safety, blood Phe concentration, PK, and immune response. Subjects | |
| | enrolled into the Substudy will also have additional PK sampling performed prior to the | |
| | dosing interruption and during the dosing interruption. To allow for PK sampling once | |
| | dosing is stopped, subjects may be admitted to a research facility within 8 hours of stopping | |
| | dosing where they will reside for at least 24 hours. After the dosing interruption, rAvPAL- | |
| | PEG administration will be re-started at the same dose level and dosing frequency that was | |
| | administered prior to the dosing interruption. Upon re-starting rAvPAL-PEG, the first dose | |
| | must be administered in the clinic and the subject must be observed for 30-60 minutes | |
| | following administration due to restarting dosing. A follow-up telephone call will be made | |
| | to the subject to monitor subject safety 24 hours following the return to dosing. Additional | |
| | PK sampling will also be performed for the first week after the dosing interruption. | |
| Section 9.1.1/Management | Subjects who qualify for self administration of study drug will be provided with | 11, 13, 21 |
| of Local and Systemic | information and instruction with regard to management of local and systemic reactions | |
| Reactions to rAvPAL-PEG | (refer to the Subject Self-Administration Training Materials). | |
| Section 9.1.1.1/Subjects | Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing | 11, 13, 21 |
| Who Have Had Previous | product that warranted early termination from PAL-002 or PAL-004 are excluded from | |
| Hypersensitivity Reactions | participation in this study. Subjects who experienced a generalized skin rash are included in | |
| to rAvPAL-PEG or a PEG- | this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in | |

| BIOM | 1ARIN° |
|------|--------|
|------|--------|


| Section No./Title | | |
|---|---|---|
| containing Product | PAL-002 or PAL-004 are eligible to participate in this study. Subjects who have had a previous reaction and are deemed eligible for participation must be premedicated orally with acetaminophen and/or antihistamines 1 hour prior to study drug dosing for the remainder of the study. The premedication dosage will be standard. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). Subjects may develop systemic, large local skin, or local skin reactions after enrollment in PAL-003. Refer to Section 9.1.1.2 for definitions of systemic and local skin reactions. For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1. | |
| Section 9.1.1.2/Definitions of Hypersensitivity Reactions to rAvPAL-PEG Administered Subcutaneously | • Skin and non-skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological; and/or a fever attributed to treatment with rAvPAL-PEG (≥ 100.4°F or ≥ 38°C). | 11, 13, 21 |
| Section 9.1.3.3.1/Local<br>Skin Reactions | Subjects who have had a local skin reaction (refer to Section 9.1.1.2 for definition) after administration of rAvPAL-PEG in PAL 001, PAL 002, or this study may continue if the symptoms do not worsen and no other symptoms have developed but may be premedicated with acetaminophen and or antihistamines (standard dosage per the package insert) 1 hour prior to the next dose of study drug dosing. Recommended premedications are | 11, 13, 21 |

| BIO | MA | R | IN° |
|-----|----|---|-----|
|-----|----|---|-----|


| Section No./Title | | |
|---|---|---|
| | acetaminophen and antihistamine (Zyrtee [cetirizine] is preferred). The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg Zyrtee or 25 to 50 mg oral Benadryl [diphenahydramine]). Because antihistamines Benadryl can cause drowsiness, it should be administered only if the subject is accompanied by a designated driver. | |
| | Symptoms of local reactions may be treated with local application of ice and non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.2.2). | |
| | If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study treatment and complete an Early Termination Visit. | |
| Figure 9.1.1.3.2/Large | Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be | 11, 13, 21 |
| Local Skin Reactions | contiguous to the rAvPAL-PEG injection site, and subjects with either type of large local skin reaction may continue dosing if the skin symptoms have resolved and no other symptoms have developed. Subjects may be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing. The location of the large local skin reaction relative to the rAvPAL PEG injection site will determine if a subject may remain in the study and continue to be administered rAvPAL PEG. An example of a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk. | |
| | Subjects who have large local skin reactions that are contiguous to the injection site may remain in the study. Subjects who have large local skin reactions that are not contiguous to the injection site may have additional assessments performed (Unscheduled | |

| BIO | M | A | R | N | 8 |
|-----|---|---|---|---|---|
|-----|---|---|---|---|---|


| Section No./Title | | |
|---|---|---|
| | Hypersensitivity Reaction Visit) per Investigator discretion and must then be terminated from the study. A decision to terminate a subject from the study must be agreed to by both the Investigator and the Sponsor's Medical Officer. | |
| Section 9.1.1.3.2.1/Large Local Skin Reactions Contiguous to Injection Site | Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may remain in the study if the skin symptoms have resolved and no other symptoms have developed. Large local skin reactions that are contiguous to the injection site should be managed as local skin reactions (refer to Section 9.1.1.3.1). For the remainder of the study, subjects must may be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to the next dose of study drug dosing. Recommended premedications are acetaminophen and antihistamine (Zyrtec [cetirizine] is preferred). The dosage will be standard (eg, 1000 mg acetaminophen and 10 mg Zyrtec or 25 to 50 mg Benadryl [diphenahydramine]). Because antihistamines Benadryl can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). | 11, 13, 21 |
| Section 9.1.1.3.2.2/Large<br>Local Skin Reactions Not<br>Contiguous to Injection<br>Site | Large local skin reactions that are not contiguous to the injection site may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure to rAvPAL-PEG and, therefore, will be managed as a systemic reaction (refer to Section 9.1.1.3.3). An example of a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk. Subjects who develop large local skin reactions that are not contiguous to the injection site after administration of rAvPAL PEG or to rAvPAL PEG or a PEG containing product may not continue to | 11, 13, 21 |

| BIO | MA | AR | IN° |
|-----|----|----|-----|
|-----|----|----|-----|


| Section No./Title | | |
|---|---|---|
| | participate in the study. Subjects may have additional assessments performed | |
| | (ie, Unscheduled Hypersensitivity Skin Reaction Visit) immediately after the reaction | |
| | (within 48 hours): serum anti-rAvPAL PEG antibodies (anti-PAL immunoglobulin G [IgG], | |
| | anti PAL immunoglobulin M [IgM], anti PEG IgG, anti PEG IgM, anti rAvPAL PEG | |
| | neutralizing antibody, and anti rAvPAL PEG immunoglobulin E [IgE]); serum tryptase | |
| | level; sedimentation rate; C reactive protein (CRP), total hemolytic complement (CH50), | |
| | and complements C <sub>1</sub> - and C <sub>4</sub> ; and clinical laboratory tests (urinalysis, chemistry, | |
| | hematology). Subjects will then be terminated from the study and should be scheduled to | |
| | complete the Early Termination Visit (refer to Section 12.4). | |
| 0.1.1.2.2/9 | | 11 12 21 |
| Section 9.1.1.3.3/Systemic | Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a definition) after | 11, 13, 21 |
| Reactions | administration of rAvPAL-PEG must stop further administrations of rAvPAL-PEG and | |
| | must immediately return to the clinic for safety assessments will be terminated from the | |
| | study. Subjects who experience generalized skin symptoms are included in this category. | |
| | Immediately after the systemic reaction (within 48 hours), subjects with generalized skin | |
| | symptoms must have additional assessments performed for safety (ie, Unscheduled | |
| | Hypersensitivity Skin Reaction Visit): serum anti-rAvPAL-PEG antibodies (anti-PAL | |
| | immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG | |
| | IgE, and anti-rAvPAL-PEG neutralizing antibody)anti PAL IgG, anti PAL IgM, anti PEG | |
| | IgG, anti PEG IgM, anti rAvPAL PEG neutralizing antibody, and anti rAvPAL PEG IgE); | |
| | serum tryptase level (optional; it is recommended that this sample be drawn immediately | |
| | after reaction); sedimentation rate; CRP, CH50, $C_1$ , $C_3$ , and $C_4$ ; skin biopsy (optional; | |
| | affected and not affected area; to be performed within 1 week of reaction); and clinical | |
| | laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1). | |
| | Following completion of the Unscheduled Systemic Reaction Visit, administration of | |

| BIOM | IAR | IN° |
|------|-----|-----|
|------|-----|-----|


| Section No./Title | |
|---|---|
| | rAvPAL-PEG may resume up to 1 week following the onset of the reaction if the systemic |
| | reaction is not IgE-mediated and the subject's safety will not be further compromised with |
| | resumed dosing. rAvPAL-PEG administration will resume at the next lowest dose level. |
| | Restarting of rAvPAL-PEG administration following a systemic reaction must be |
| | performed in the clinic for the first week of resumed dosing. Subjects must be premedicated |
| | orally with acetaminophen and/or antihistamines (standard dosage per the package insert) |
| | 1 hour prior to study drug dosing for the remainder of the study. Additionally, subjects must |
| | be closely monitored for 30-60 minutes following every administration of study drug. |
| | Because antihistamines may cause drowsiness, the subject must be accompanied by a |
| | designated driver (if applicable). |
| | If blood Phe concentrations are not 60-600 μmol/L following 1 week of daily |
| | administration at the lowered dose cohort and there is no further evidence of toxicity (ie, |
| | another systemic reaction attributed to rAvPAL-PEG administration or clinically significant |
| | abnormal laboratory test results), the subject may be administered the next highest dose |
| | level in the clinic per the allowable dose increases outlined in Section 9.1.2. Subjects must |
| | be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the |
| | package insert) 1 hour prior to study drug dosing for the remainder of the study. |
| | Additionally, subjects must be closely monitored for 30-60 minutes following every study |
| | drug administration. Because antihistamines may cause drowsiness, the subject must be |
| | accompanied by a designated driver (if applicable). |
| | Subjects who have a systemic reaction without generalized skin symptoms may have these |
| | assessments performed per Investigator discretion. Subjects will then be terminated from |
| | the study and should be scheduled to complete the Early Termination Visit (refer to |
| | Section 12.4). |




| Section No./Title | | |
|---|---|---|
| Section 9.1.2/Dose<br>Modifications | After any modifications (increases or decreases) to dose level or frequency, subjects should remain in the clinic for observation for at least 2 hours following the injection of study drug. The Investigator should remain at the site to assess the subject for safety. | 2, 3, 21, 22, 23 |
| Section 9.1.2.1/Dose Increase Methodology | Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Study Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations. Blood Phe levels will be measured 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed. For subjects from PAL-002Depending upon the response to rAvPAL-PEG in PAL-002, an individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows. • The dose may be increased by increments of no more than 10-fold higher than the subject's current dose. • When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, and 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg) that were defined in the previous study (PAL-002)-or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 µmol/L) and drug concentrations, as well as any adverse events (any hypersensitivity reaction) for an individual subject. • The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed \$\frac{5}{2}.0 \text{ mg/kg}, including subjects who receive more than 1 dose/week. Subjects who increase their dose frequency should perform the Interim Dosing Visit assessments (refer to Section 12.3.6\frac{5}{2} \text{ and Table 2.1.3} and Table 2.1.4 Table 2.1.4 to ). | 2, 3, 21, 22, 23 |

| BIO | M | A | R | N | 8 |
|-----|---|---|---|---|---|
|-----|---|---|---|---|---|


| Section No./Title | | |
|---|---|---|
| | <ul> <li>When a dose is increased (either by increasing the dose level or by increasing the frequency of dosing), the subject must remain in the clinic be observed for a minimum of 30-60 minutes hours following the first modified dose administration, and an Investigator will remain on site during this time. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.</li> <li>Only 1 dose (level or frequency) adjustment is allowed every 2 weeks.</li> <li>Blood Phe levels will be measured daily for 3 days after each dose increase (fingerstick is acceptable); more frequent or daily blood Phe measurements may be performed.</li> </ul> | |
| Section 9.1.2.2/Dose Decrease Methodology | A subject's diet should be assessed prior to any dose decreases. Changes to diet should only be made if a subject's blood Phe concentrations < 120 μmol/L. If a subject's blood Phe level is < 120 μmol/L, the subject's dietary Phe intake should be increased to achieve a stable blood Phe concentration of 120 600 μmol/L. If the subject's blood Phe level is < 120 μmol/L despite a high Phe diet, the rAvPAL PEG dose will then be decreased. The subject will be asked about any changes to diet prior to any dose adjustments, and any changes to diet should be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. | 2, 3, 21, 22, 23 |
| | All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 µmol/L> 30% change from baseline) and drug concentrations, as well as any adverse eventstoxicity (any hypersensitivity reaction as defined in Section 9.1.1.2). Dose decreases may occur for safety (ie, blood Phe concentration < 120 µmol/L) or other toxicityany adverse event that may be improved with a lower, more frequent dose). | |
| | A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between | |

**B**OMARIN

PAL-003


| Section No./Title | | |
|---|---|---|
| | these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced. | |
| Section 9.1.3/ <u>Safety</u> <u>Assessment</u> Stopping Criteria | If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principle Investigator (PI) and the Study Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level. | 8 |
| Section 9.1.4/ <u>Stopping</u> <u>Criteria</u> | Ifn addition, if 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will be evaluated and halted and no subject will be treated at a higher dose level until a safety assessment will be is completed. In addition, the Food and Drug Administration (FDA) may will be notified of this occurrence if appropriate. | 8 |
| Section 9.3.1/Inclusion<br>Criteria | Individuals eligible to participate in this study must meet all of the following criteria: 1. Must have completed participation and all protocol-defined study drug in PAL-002 or PAL-004. | 4 |
| Section 9.3.2/Exclusion<br>Criteria | Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study: 1. Use of any investigational product (with the exception of rAvPAL-PEG) or | 4, 11 |
| BIO | MA | ٩R | IN. |
|-----|----|----|-----|
|-----|----|----|-----|


| Section No./Title | | |
|---|---|---|
| | investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments. | |
| | 2. Use of any medication <u>other than rAvPAL-PEG</u> that is intended to treat PKU within 14 days prior to the administration of study drug. | |
| | 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation. | |
| | <ol> <li>A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.</li> <li>Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL-002 or PAL-004.</li> </ol> | |
| Section 9.3.3/Removal of<br>Subjects from Treatment or<br>Assessment | Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study treatment should continue to perform the study tests and evaluations until study completion. For subjects who | 8, 27 |
| | discontinue from the study, the tests and evaluations listed for the Early Termination Visit | |




| Section No./Title | | |
|---|---|---|
| | should be carried out (refer to Section 12.4). | |
| | BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance. | |
| | Reasons for which the Investigator or BioMarin may withdraw a subject from the study treatment include, but are not limited to, the following: | |
| | • Subject experiences a serious or intolerable adverse event (AE). | |
| | <ul> <li>Subject develops a clinically significant laboratory abnormality.</li> </ul> | |
| | <ul> <li>Subject requires medication prohibited by the protocol.</li> </ul> | |
| | <ul> <li>Subject becomes pregnant (refer to Section 10.3 for details on the reporting<br/>procedures to follow in the event of pregnancy).</li> </ul> | |
| | Reasons for which the Investigator or BioMarin may withdraw a subject from the study | |
| | include, but are not limited to, the following: | |
| | <ul> <li>Subject does not adhere to study requirements specified in the protocol.</li> </ul> | |
| | • Subject was erroneously admitted into the study or does not meet entry criteria. | |
| | • Subject is lost to follow-up. | |
| | <ul> <li>Subject becomes pregnant (refer to Section 10.3 for details on the reporting<br/>procedures to follow in the event of pregnancy).</li> </ul> | |
| Section 9.3.4/Subject | Subjects will retain the same subject number assigned in PAL-002 or PAL-004. | 4 |
| Identification and | | |




| Section No./Title | | |
|---|---|---|
| Replacement of Subjects | | |
| Section 9. 4/Treatments | Upon enrollment into this study, subjects from PAL-002 will be dosed with the same or higher dose that was administered upon completion of PAL-002. Subjects enrolling from PAL-004, will be administered the same dose that was administered upon completion of PAL-004. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on on available information regarding a subject's blood Phe level (60-600 μmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600 μmol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed to by the PI and the Study Medical Officer, based upon the subject's response to doses. Subjects may self administer study drug at home if approved by the Sponsor's Medical Officer and if adequate training is provided. Subjects may be eligible to self administer study drug if he or she meets the following criteria: • The subject has not experienced any CTCAE Grade 3 or higher adverse event. • The subject has not experienced any hypersensitivity reaction to rAvPAL-PEG for at least 4 weeks. • The subject has no cognitive impairments that may increase the safety risk of self administration per the assessment of the PI. | 10 |

| BIO | MA | AR | IN° |
|-----|----|----|-----|
|-----|----|----|-----|


| Section No./Title | |
|---|---|
| | Sponsor's Medical Officer. |
| | The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely. |
| | The subject has been provided with epinephrine and has been trained on when and how to administer it. |
| | Qualified study site personnel will train each eligible subject on all procedures for self |
| | administration of study drug under the supervision of the PI. Qualified study site personnel |
| | will also be required to observe the subject prepare and perform at least 1 injection prior to |
| | allowing the subject to self administer a dose at home. The patient will see a study site |
| | nurse or home healthcare nurse in person every week to ensure that the subject continues to |
| | perform all self-administration procedures correctly, to assess for adverse events, and to |
| | answer questions throughout the duration of the study. The study site nurse or home |
| | healthcare nurse will also perform the regularly scheduled assessments and procedures as |
| | outlined in Table 2.1.1 and Section 12; the subject must perform a clinic visit monthly at |
| | minimum. Training materials and other information specific to the study site personnel are |
| | provided in the Subject Self-Administration Training Materials. |
| | Subjects who are eligible for self administration will be provided with a Subject Study |
| | Manual, Self-administration training materials will be provided in the Subject Study |
| | Manual to supplement the in-person training provided by the qualified study site personnel. |
| | The Subject Study Manual will include step-by-step instruction on the following: |
| | How to prepare and perform the injections of study drug safely. |
| | How to receive, track, store, prepare, and return both used and unused study drug. |




| Section No./Title | | |
|---|---|---|
| | <ul> <li>How to safely use and dispose of syringes used for injections of study drug.</li> <li>How to care for their injection site after an injection of study drug.</li> <li>How to identify an adverse reaction and how to report this reaction to the study site.</li> <li>How and when to use epinephrine.</li> <li>Who to contact at the study site in case of an emergency.</li> </ul> The PI or the Sponsor's Medical Officer may request that self administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse. | |
| Section 9.4.1/Treatments Administered | BioMarin and/or its designee will provide the study site with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplyingthe study drug to subjects who qualify for self administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites. Information regarding supplying study drug to subjects who qualify for self administration is provided in the Subject Self-Administration Training Materials. | 10, 27 |
| Section 9.4.3/Storage | At the study site, all IP must be stored at $5 \pm 3^{\circ}$ C ( $41 \pm 5^{\circ}$ F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures. | 10, 27 |




| Section No./Title | | |
|---|---|---|
| | Specific instructions for storage of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials. | |
| Section 9.4.4/Directions for Administration | Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.02 mg/kg. Information for subjects who are participating in the Substudy and re-start rAvPAL-PEG dosing is provided in Section 9.1. Information for dosing of subjects who enroll into this study after completing Study PAL-004 is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10. Instructions for administration of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency maywill need to be re-evaluated (refer to Section 9.4.10). | 2, 10, 27 |
| Section 9.4.5/Method of<br>Assigning Subjects to<br>Treatment Groups | Subjects will retain the same subject number used in PAL-002 or PAL-004. | 4, 27 |

| BIO | MA | RI | N° |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| Section 9.4.6/Selection of Doses Used in the Study | This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 6120-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study and the ongoing study, PAL-002, to date (JAN2011). The doses for this study are based upon the results of nonclinical studies and PAL 001. The no observable adverse effect level (NOAELs) from nonclinical studies in rats and monkeys represents a greater than 100 fold safety factor over the starting dose administered in PAL 002 (0.001 mg/kg). | 3 |
| Section 9.4.6.1/Selection<br>of Timing of Dose for<br>Each Subject | Study drug will be administered in the morning by clinic staff or other qualified and trained study personnel. Subjects may self administer study drug at home if approved by the Sponsor's Medical Officer and if adequate training is provided (refer to Section 9.4). | 19 |
| Section 9.4.8/Prior and Concomitant Medications | Use of any investigational product (with the exception of rAvPAL-PEG used in PAL-002 or PAL-004) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior local skin reaction to rAvPAL-PEG or a | 4, 11 |

| BIO | M | A | R | IN° |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | | |
|---|---|---|
| | PEG-containing product will be premedicated with acetaminophen and/or antihistamines (refer to Section 9.1.1). If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Study Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit. Subjects who have had a prior systemic reaction to rAvPAL-PEG or a PEG-containing product are excluded frommay participateion in this study (refer to Section 9.1.1). | |
| Section 9.4.10/Dose Interruption and Missed Doses | Information for subjects who are participating in the Substudy and re-start rAvPAL-PEG dosing is provided in Section 9.1. Information for dosing of subjects who enroll into this study after completing Study PAL-002 or Study PAL-004 is provided in Section 9.1. During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator in consultation with the Sponsor's Medical Officer. Subjects who miss more than 2 consecutive weekly doses (weekly dosing schedule) or 3 consecutive daily doses (daily dosing schedule) for whatever reason may continue participation in this study. After a dosing interruption, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects should continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 2.1.1, Table 2.1.2, Table 2.1.3, and Table 2.1.4) during any dosing interruption. | 7 |




| Section No./Title | | |
|---|---|---|
| | Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study treatment per discretion of the Sponsor or Investigator (refer to Section 9.3.3). | |
| Section 9.5/Investigational Product Accountability | The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), <u>IP returned</u> , and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data. | 27 |
| Section 9.5.1/Return and Disposition of Clinical Supplies | Subjects who qualify for self administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials). | 10 |
| Section 9.6/Dietary or Other Protocol Restrictions | Subjects will be instructed that diet should not be altered during the course of the study-except as necessary for safety. If a subject's blood Phe concentration is < 120 µmol/L, the subject's diet will be adjusted to maintain blood Phe concentrations of 120 600 µmol/L. Changes to diet will be made per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigaor in consultation with the Sponsor's Medical Officer. A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next dose of study drug. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4. | 6 |

| BIO | MA | RI | N° |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| Section 9.7.1.5/Chest X-Ray | A chest X-ray will be performed at the <u>Screening</u> , Month 12, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health. | 24 |
| Section 9.7.2.1/Blood Phenylalanine Concentrations | Blood samples for Phe concentration measurements will be drawn in the morning, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 2.1.1, Table 2.1.2, Table 2.1.3, and Table 2.1.4). In addition, after each administration of study drug, the subject will have a blood Phe measurement by fingerstick as outlined in Table 2.1.1, Table 2.1.2, Table 2.1.3, and Table 2.1.4. This may be done by the subject at home. Subjects who have their dose frequency increased will have additional Phe assessments performed as outlined in Table 2.1.3: and Table 2.1.4: | 19, 27 |
| Section<br>9.7.3/Pharmacokinetic<br>Variables | Steady state PK (predose samples) of rAvPAL PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentration (120 600 µmol/L) for a minimum of 2 weeks (to allow assessment of blood Phe concentrations) and no further dose modification is planned. Once this target has been achieved, PK samples will be collected predose on the same day each week for 3 consecutive weeks. Subjects enrolled in the Substudy will have additional PK sampling performed prior to the planned dosing interruption and upon re-introduction of rAvPAL-PEG. For subjects participating in the Substudy, PK sampling will be performed as follows: | 1, 14 |

| BIO | M | A | R | IN |
|-----|---|---|---|----|
|-----|---|---|---|----|


| Section No./Title | | |
|---|---|---|
| | <ul> <li>When dosing is stopped, PK sampling will be performed prior to the final dose and then postdose at 8 hours, 12 hours, 16, hours, 24 hours, 48, hours, 72 hours, 96 hours, 144 hours, 168 hours, and 216 hours.</li> <li>When dosing is re-started, PK sampling will be performed predose and then postdose at 24 hours, 48 hours, 72 hours, 120 hours, and 168 hours.</li> </ul> | |
| | Subjects who have increased their dose frequency to twice weekly or daily will have addition PK assessments performed for 5 weeks after the change in dose regimen (refer to Section 12.3.5 and Table 2.1.3: -and Table 2.1.4: ). BioMarin will perform the analysis. | |
| Section 9.7.4/Exploratory Efficacy Variable | Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each week. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator. | 5 |
| Section 9.7.5.2/Antibody Testing | Immunogenicity will be assessed by determining antibody immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1.3.3).1) anti-rAvPAL immunoglobulin G (IgG) antibodies, 2) anti-rAvPAL immunoglobulin M (IgM) antibodies, 3) anti-PEG IgG antibodies, 4) anti-PEG IgM antibodies, 5) anti-rAvPAL PEG immunoglobulin E (IgE) antibodies, and 6) anti-rAvPAL PEG Enzyme Activity Neutralizing antibodies (NAb), and 7) rAvPAL | 23, 27 |




| Section No./Title | | |
|---|---|---|
| | PEG antibody clearing complexes (if needed). Validated immunogenicity assays will be used per the time points indicated in the Schedule of Events (Table 2.1.1 and Table 2.1.2). BioMarin will perform the analysis except for anti rAvPAL PEG IgE antibodies, which will be assessed by a Contract Research Organization. | |
| Section 9.7.6/Clninical<br>Laboratory Assessments | All clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not any abnormal the result is clinically significant. Table 9.7.6.1: Clinical Laboratory Tests has been revised to include information for subjects who have a positive result from the urine pregnancy test. | 27 |
| Section 10.1/ Adverse Events | According to the ICH definition, an AE (or adverse experience) is "any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the IP." For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a patient administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following: AEs not previously observed in the subject that emerge during the course of the study. Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study. Complications that occur as a result of non-drug protocol-imposed interventions | 15 |
| | • Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment run- | |

| B <sub>2</sub> OI | MA | RI | N° |
|-------------------|----|----|----|
|-------------------|----|----|----|


| Section No./Title | |
|---|---|
| | in). |
| | An adverse drug reaction (ADR) is described by the ICH as "all noxious and unintended |
| | responses to a medicinal product related to any dose." This means that a causal relationship |
| | between a medicinal product and an AE is at least a reasonable possibility, ie, the |
| | relationship cannot be ruled out An adverse drug reaction is any AE for which there is a |
| | reasonable possibility that the study drug caused the AE. "Reasonable possibility" means |
| | there is evidence to suggest a causal relationship between the study-drug and the AE. |
| | An AE may include intercurrent illnesses or injuries that represent an exacerbation (increase |
| | in frequency, severity, or specificity) of pre existing conditions (eg, worsening of asthma). |
| | Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series |
| | of terms relating to a diagnosis. |
| | The reporting period for non serious AEs is the period from the first administration of study |
| | drug through the final F/U Visit or at the ETV. If a non-serious AE remains unresolved at |
| | the conclusion of the study, the PI and medical monitor will make a joint clinical |
| | assessment as to whether continued follow up of the AE is warranted, and the results of this |
| | assessment must be documented. Resolution is defined as the return to baseline status or |
| | stabilization of the condition with the expectation that it will remain chronic. |
| | The study period during which all non-serious AEs and SAEs will be reported begins after |
| | informed consent is obtained and the first adminstration of study drug and continues until |
| | 4 weeks following the last administration of study drug or the last visit of the treatment |
| | period (refer to Section 12). After informed consent but prior to initiation of study |
| | treatment, only SAEs associated with any protocol-imposed interventions will be reported. |
| | The criteria for determining, and the reporting of SAEs is provided in The Investigator will |
| | assess AEs for severity, for relationship to IP, and as to whether the event meets one or |
| | more of the definitions of a serious adverse event (SAE; refer to Section 10.2). |




| Castian No /Title | | | | |
|---|---|---|---|---|
| Section No./Title | | | | |
| | The Investigator s | The Investigator should follow all unresolved AEs until the events are resolved or | | |
| | stabilized, the sub | stabilized, the subject is lost to follow-up, or it has been determined that the study treatment | | |
| | or study participation is not the cause of the AE. Resolution of AEs (with dates) should be | | | |
| | documented on the appropriate CRF page(s) and in the subject's medical record. | | | |
| | The Investigator responsible for the care of the patient or qualified designee will assess AEs | | | |
| | for severity, relati | ionship | to study-drug, and seriousness (see Section 10.2 for SA | <u>AE</u> |
| | definition). Sever | ity (as i | n mild, moderate or severe headache) is not equivalent | to |
| | seriousness, which | h is bas | ed on patient/event outcome or action criteria usually a | ssociated |
| | with events that p | ose a th | reat to a patient's life or functioning. Seriousness (not | severity) |
| | | | ning regulatory reporting obligations. | |
| | The Investigator y | will dete | ermine the severity of each AE <u>using the National Can</u> | cer Institute |
| | - | | logy Criteria for Adverse Events (CTCAE) v4. Advers | |
| | | | ing CTCAE term will be assessed according to the gen | |
| | guidelines for grading used in the CTCAE v4 as stated below.and will record it on the | | | |
| | source documents and AE CRF, using the CTCAE v 3 grades defined below. Events that | | | |
| | | | 5 are serious events and require completion of both an | |
| | and AE eCRF. | | 1 | |
| | Gra | ade | Description | |
| | 1 Mild: asymptomatic or mild symptoms; clinical or | | | |
| | diagnostic observations only; intervention not | | | |
| | | | indicated | |
| | 2 | | Moderate: minimal, local or noninvasive | |
| | | | intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> | |
| | | | instrumental activities of daily fiving (ADL) | |




| Section No./Title | | |
|---|---|---|
| | Severe or medically significant but not immediately life-threatening: hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL) | |
| | 4 Life threatening or debilitating: consequences; urgent intervention indicated <sup>b</sup> | |
| | 5 Death related to AE | |
| | Grade 4 and 5 AEs should always be reported as SAEs. | |
| | <sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for | |
| | groceries or clothes, using the telephone, managing money. | |
| | <sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding | |
| | oneself, using the toilet, taking medications, not bedridden. | |
| | The term "severe" is often used to describe the intensity (severity) of a specific event (as in | |
| | mild, moderate, or severe myocardial infarction); the event itself, however, may be of | |
| | relatively minor medical significance (such as severe headache). This is not the same as | |
| | "serious," which is based on subject/event outcome or action criteria usually associated | |
| | with events that pose a threat to a subject's life or functioning. Seriousness (not severity) | |
| | serves as a guide for defining regulatory reporting obligations. | |
| | The Investigator will determine the relationship of an AE to the <u>Hestudy drug</u> and will | |
| | record it on the source documents and AE CRF, using the categories defined below. | |
| Section 10.2/Serious | A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 | 15 |
| Adverse Events | or more of the following criteria: | |




| Section No./Title | |
|---|---|
| | Is fatal. |
| | <u>Is life threatening.</u> |
| | Note: Life-threatening refers to an event that places the patient at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death. |
| | Requires or prolongs inpatient hospitalization. |
| | Results in persistent or significant disability or incapacity. |
| | Is a congenital anomaly or birth defect in the child or fetus of a patient exposed to IP prior to conception or during pregnancy. |
| | Is an important medical event or reaction. |
| | A SAE is defined as any AE that: |
| | • Results in death. |
| | • Is life threatening, that is, places the subject at immediate risk of death from the event as it occurred. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death. |
| | <ul> <li>Requires in patient hospitalization or prolongation of an existing in patient hospitalization. Admission of a subject to the hospital as an in patient as a result of an AE, even if the subject is released on the same day, qualifies as hospitalization.</li> </ul> |
| | <ul> <li>Results in persistent or significant disability or incapacity. An event qualifies as resulting in a persistent or significant disability or incapacity if it involves a substantial disruption of the subject's ability to carry out usual life functions. This definition is not intended to include experiences of relatively minor or temporary medical significance.</li> </ul> |
| | <ul> <li>Is a congenital anomaly or birth defect, that is, an AE that occurs in the child or<br/>fetus of a subject exposed to IP prior to conception or during pregnancy.</li> </ul> |

| BIO | M | A | R | IN |
|-----|---|---|---|----|
|-----|---|---|---|----|


| Section No./Title | |
|---|---|
| | • Is an important medical event that does not meet any of the above criteria, but may jeopardize the subject or require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such events are intensive treatment in the emergency room, allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse. |
| | More than one of the above criteria may apply to any specific event. |
| | The reporting period for SAEs begins after informed consent is obtained, and continues until 4 weeks following the last administration of study drug or End of Treatment Visit. The reporting period for SAEs begins earlier than non serious AEs and is the period from the time of signing of the ICF-through 4 weeks after the last dose or at the ETV. SAEs reported to the Investigator outside of this reporting period will be reported to BioMarin if, in good medical judgment, the event has any bearing on the study data. SAEs must be followed by the Investigator until resolution, even if this extends beyond the study reporting period. Resolution of an SAE is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic. |
| | Any SAE, whether or not considered related to study drug, will be reported immediately |
| | (within 24 hours) to BioMarin Pharmacovigilance by fax using the study specific |
| | SAE Report Form. In addition to the outcome of the SAE, any medication or other |
| | therapeutic measures used to treat the event will be recorded on the appropriate CRF |
| | page(s). Investigators should not wait to collect additional information that fully documents |
| | the event before notifying BioMarin Pharmacovigilance of an SAE. BioMarin may be |
| | required to report certain SAEs to regulatory authorities within 7 calendar days of being |
| | notified about the event; therefore, it is important that Investigators submit additional |
| | information requested by BioMarin as soon as it becomes available. All SAEs, whether or |
| | not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form to BioMarin |

| B <sub>2</sub> OI | MA | RI | N° |
|-------------------|----|----|----|
|-------------------|----|----|----|


| Section No./Title | |
|---|---|
| | Pharmacovigilance (BPV). ). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the patient's medical record. |
| | For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report). At the last scheduled visit, the Investigator should instruct each subject to report any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study treatment. |
| | The investigator should notify the study Sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior study treatment. The Sponsor should also be notified if the Investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that participated in this study. |

| BIO | M | A | R | N | 8 |
|-----|---|---|---|---|---|
|-----|---|---|---|---|---|


| Section No./Title | | |
|---|---|---|
| Section 10.3/Pregnancy | Pregnancy in a subject or partner should be reported immediately (within 24 hours of the site becoming aware of the pregnancy) to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up Form in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information. | 15 |
| Section 10.4/Urgent Safety Measures | The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours. Examples of situations that may require urgent safety measures include discovery of the | 15 |

**B**OMARIN

PAL-003


| Section No./Title | | |
|---|---|---|
| | <ul> <li><u>Immediate need to revise the IP administration (ie, modified dose amount or frequency not defined in protocol).</u></li> <li><u>Lack of study scientific value, or detrimental study conduct or management.</u></li> <li><u>Discovery that the quality or safety of the IP does not meet established safety requirements.</u></li> </ul> | |
| Section 11.2/Diet Diary | A 3-day diet diary will be issued to subjects for completion and will be brought to each clinic visit for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6. | 5 |
| Section 12.2/Screening<br>Visit | • <u>Chest X-ray</u> For subjects who participated in PAL-002 <u>or PAL-004</u> , these assessments may be the same <u>as those</u> used for the Week 16 Visit of PAL-002 <u>or the Week 16 visit of PAL-004</u> , if they occur within 28 days from Day 1. | 24, 26 |
| Section 12.3/Treatment<br>Period | During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done | 26 |

| BIO | MA | RI | N° |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| | predose unless otherwise specified. <u>Subjects must have AEs and concomitant medications</u> <u>assessed and an injection-site inspection performed whenever dose is administered even if</u> <u>the administration does not coincide with a scheduled clinic visit.</u> | |
| | If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done on the third daydaily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment. | |
| Section 12.3.1/Day 1 (Week 1) | <ul> <li>3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.)</li> <li>Predose PK sample</li> <li>Predose bBlood Phe and plasma tyrosine concentration</li> <li>Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies) (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-PAL PEG neutralizing antibody, and anti-rAvPAL PEG IgE)</li> <li>Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)</li> <li>For subjects enrolling into this study from Study PAL-004, first dose of rAvPAl-pEG must be given in the clinic setting and a telephone follow-up with the subject must be performed 24 hours later to assess safety issues.</li> </ul> | 26 |

| BIO | M | A | R | IN | 8 |
|-----|---|---|---|----|---|
|-----|---|---|---|----|---|


| Section No./Title | | |
|---|---|---|
| Section 12.3.2/Weekly | Weekly visits do not require an in-clinic visit if conducted by a home healthcare | 26 |
| Visits | professional. However, dose modifications must be peformed in the clinic. Subjects must | |
| | have AEs and concomitant medications assessed and an injection-site inspection performed | |
| | whenever dose is administered even if the administration does not coincide with a | |
| | scheduled clinic visit. | |
| | Predose-PK sample | |
| | o For subjects participating in the Substudy, refer to Section 12.3.3. | |
| | OPER investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120 600 μmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2 3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes. | |
| | Predose bBlood Phe and plasma tyrosine concentration | |
| | Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120 600 μmol/L for the majority of the 3 months), the predose plasma Phe and tyrosine assessments may be skipped at the weekly visits and performed at the monthly visits for the first year then 2-3 months thereafter. The weekly plasma Phe assessment may be replaced with a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes. | |
| | <ul> <li>Administer study drug (study drug may be administered on additional days during<br/>the week as determined by the Investigator, in agreement with the Study Medical<br/>Officer)</li> </ul> | |
| | o For subjects participating in the Substudy, refer to Section 12.3.3. | |




| Section No./Title | | |
|---|---|---|
| Section 12.3.3/Substudy | The following study activities will be performed on Day 1 of the Substudy (ie, final dose | 1, 26 |
| Visits (Weekly) | prior to interruption), Day 8, Day 15, Day 22, and Day 29 (ie, restart administration of | |
| | study drug) for subjects participating in the Substudy: | |
| | Physical examination | |
| | Vital signs, including weight | |
| | Clinical laboratory tests | |
| | Sedimentation rate | |
| | Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) | |
| | <ul> <li>Injection-site inspection (predose; postdose on Day 1; during weekly visit on Day 8, 15, 22; and postdose on Day 29)</li> </ul> | |
| | Assessment of AEs | |
| | Concomitant medications | |
| | • <u>Diet query</u> | |
| | • 3-day diet diary | |
| | • Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies,) | |
| | Blood Phe and plasma tyrosine concentration | |
| | <ul> <li>When dosing is stopped, sampling for blood Phe assessment only will</li> </ul> | |
| | be performed prior to the final dose and then postdose at 8 hours, 12 | |
| | hours, 16 hours, 24 hours, 48, hours, 72 hours, 96 hours, 144 hours, | |
| | 168 hours, and 216 hours. | |
| | When dosing is re-started, sampling for blood Phe assessment only will | |

| BIO | M | A | R | IN° |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | | |
|---|---|---|
| | be performed predose and then postdose at 24 hours, 48 hours, 72 hours, 120 hours, and 168 hours. • PK sample • For subjects participating in the Substudy, additional PK sampling will be performed upon the final dose prior to the planned dosing interruption and upon re-introduction of rAvPAL-PEG. Refer to Section 9.7.3 • Administer study drug (Day 29 only) • For subjects participating in the Substudy, administration of rAvPAL-PEG will not be performed for approximately 4 consecutive weeks regardless of their dosing regimen (dose level and frequency). After approximately 4 weeks of no dosing, rAvPAL-PEG administration will be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of readministration must be given in the clinic setting, and a telephone follow-up with the subject must be performed 24 hours later to assess safety issues. | |
| Section 12.3.4/Monthly<br>Visits (Week 4, 8, 12, etc) | Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. Monthly visits consist of all weekly activities and include additional activities and must be performed in the clinic. The following study activities will be performed at the monthly visits beginning with Week 4: | 26 |
| | • Predose-PK sample (subjects who are on a stable dosing regimen for ≥ 3 months | |




| Section No./Title | |
|---|---|
| | only) |
| | <ul> <li>For subjects participating in the Substudy, refer to Section 12.3.3.</li> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120 600 μmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2 3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.</li> </ul> |
| | Predose bBlood Phe and plasma tyrosine concentration |
| | O Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120 600 μmol/L for the majority of the 3 months), the predose plasma Phe and tyrosine assessments may be skipped at the weekly visits and performed at the monthly visits for the first year then 2 3 months thereafter. The weekly plasma Phe assessment may be replaced with a Phe fingerstick test. Weekly testing should resume if the subject's dosing regimen changes. |
| | <ul> <li>Serum <u>anti-rAvPAL-PEG</u> antibodies (<u>anti-PAL IgG</u>, <u>anti-PAL IgM</u>, <u>anti-PEG IgG</u>, <u>anti-PEG IgM</u>, <u>and anti-rAvPAL-PEG neutralizing antibodies</u>) (<del>anti-PAL IgG</del>, <u>anti-PAL IgM</u>, <u>anti-PEG IgG</u>, <u>anti-PAL IgM</u>, <u>anti-PEG IgM</u>, <u>anti-rAvPAL PEG neutralizing antibody</u>, <u>and anti-rAvPAL PEG IgE</u>)</li> </ul> |
| | Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer) |
| | o For subjects participating in the Substudy, refer to Section 12.3.3. |

| BIO | M | A | R | IN° |
|-----|---|---|---|-----|
|-----|---|---|---|-----|


| Section No./Title | | |
|---|---|---|
| Section 12.3.5/Quarterly<br>Visits (Week 12, 24, 36,<br>etc) | Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. | 26 |
| | <ul> <li>Predose PK sample (subjects who are on a stable dosing regimen for ≥ 3 months only)</li> <li>For subjects participating in the Substudy, refer to Section 12.3.3.</li> <li>Per investigator discretion, once a subject is on a stable dosing regimen for at least 3 months (as evidenced by blood Phe levels of 120 600 µmol/L for the majority of the 3 months), the predose PK assessment may be skipped at the weekly visits and performed at the monthly visits for the first year then 2 3 months thereafter. Weekly sampling should resume if the subject's dosing regimen changes.</li> </ul> | |
| | <ul> <li>Predose bBlood Phe and plasma tyrosine concentration</li> <li>Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies) (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL PEG neutralizing antibody, and anti-rAvPAL PEG IgE)</li> </ul> | |
| | <ul> <li>Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Study Medical Officer)</li> <li>For subjects participating in the Substudy, refer to Section 12.3.3.</li> </ul> | |
| Section 12.3. <u>6</u> 5/Interim Dosing Visit | Subjects increase their dose frequency to 2x/week will have an additional predose PK sample obtained prior to administration of the first 4 doses (ie, for 2 weeks after the dose frequency increase). For the remaining 3 weeks after | 26 |

| BIO | M | A | R | IN |
|-----|---|---|---|----|
|-----|---|---|---|----|


| Section No./Title | | |
|---|---|---|
| | the dose frequency increase, a PK sample will be obtained weekly prior to the first dose. Refer to Table 2.1.3: for the Interim Dosing Visit schedule. Subjects who have their dose frequency increased to daily will have additional PK samples obtained every day for the first week: 12 hours after the first daily dose and predose every day for the rest of the week. After the first week of daily dosing, subjects will have weekly PK samples obtained for 4 additional weeks. Refer to Table 2.1.4: for the Interim Dosing Visit schedule. | |
| Section 12.3.7/Unscheduled Hypersensitivity Reaction Visit | Subjects who have a systemic reaction, including a generalized skin reaction, or a large local skin reaction that is not contiguous to the injection site after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 48 hours) the reaction. Subjects who have other systemic symptoms or a large local skin reaction that is not contiguous to the injection site (refer to Section 9.1.1) may have these assessments performed per investigator discretion. • CRP, CH50, C1, C3, and C4 • Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies) (anti PAL IgG, anti PAL IgM, anti PEG IgG, anti PEG IgM, anti-rAvPAL PEG neutralizing antibody, and anti rAvPAL PEG IgE) • Serum tryptase level • Perform immediately after reaction if possible. • Assessment is optional for subjects who have a generalized skin reaction per investigator discretion. • Skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction) | 11, 21, 26 |

| BIO | MA | ٩R | IN |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| Section 12.4/Early | Following completion of the Unscheduled Hypersensitivity Reaction Visit assessments, the subject may resume treatment with study drug per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. Subjects who have had an IgE-mediated reaction must be discontinued from further study drug administration. Subjects who do not have an IgE-mediated reaction may resume study drug administration under close monitoring; subjects must be premedicated orally with acetaminophen and/or antihistamines 1 hour prior to study drug dosing for the remainder of the study (refer to Section 9.1.5.3.3). Subjects should then return to the clinic 4 weeks after their last dose of rAvPAL PEG for the Early Termination Visit assessments (refer to Section 12.4). The Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug. | 26 |
| Termination Visit | Subjects who terminate from study treatment early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion. Subjects who complete an Unscheduled Hypersensitivity Reaction Visit (refer to Section 12.3.6) will be terminated from the study. Subjects will then return 4 weeks after the last dose of study drug for the Early Termination Visit. • 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.) • Serum anti-ravPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PAL IgM, anti-PEG IgG, anti-PAL IgM, anti-PEG IgG, anti-PAL IgM, anti-PAL IgM | |

| BIO | MA | AR | IN |
|-----|----|----|----|
|-----|----|----|----|


| Section No./Title | | |
|---|---|---|
| Section 12.5/Final Follow-<br>up Visit | <ul> <li>3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Final Follow-up Visit.)</li> <li>Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies) (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PAL IgM, anti-rAvPAL PEG IgE)</li> </ul> | 26 |
| Section 14.2/Safety<br>Analysis | All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by—subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Safety will be evaluated on the incidence of AEs, including serious AEs (SAEs), and clinically significant changes in vital signs and laboratory test results. Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, ECG results, and X-ray results will also be provided. The verbatim terms reported on CRFs to identify AEs will be coded using MedDRA. Treatment emergent AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. Changes from baseline in vital signs and laboratory test results will be summarized with descriptive statistics. | 26 |

**B**IOMARIN

PAL-003


| Section No./Title | | |
|---|---|---|
| Section 14.3/Pharmacokinetic | Data from all subjects who complete at least 2 weeks of the study will be included in the PK analysis. | 1 |
| Analysis | Steady state PK (predose samples) of rAvPAL PEG will be evaluated in PKU subjects after the subject has achieved and maintained target blood Phe concentrations (120 <u>60</u> 600 µmol/L) for a minimum of 2 weeks and no further dose modification is planned. | |
| | Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration $(T_{max})$ , maximum plasma concentration $(C_{max})$ , half life $(t_{1/2})$ , and clearance $(CL/F)$ . | |
| | Should data become available from PAL-002 or PAL-004 that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the Sponsor's | |
| | Medical Officerbut not to exceed 3x/week. | |
| Section 14.4/ Efficacy<br>Analysis | Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis. | 1, 3, 5 |
| | Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 12060-600 µmol/L will be summarized by each scheduled time point. | |
| | The relationship of dietary Phe intake (per information reported on the subject diet diary) | |




| Section No./Title | | |
|---|---|---|
| | and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis. Information regarding this exploratory analysis will be provided in the Statistical Analysis Plan. For subjects who completed the Substudy, the effect of stopping and re-starting rAvPAL-PEG dosing on safety, blood Phe level, and immune response will be explored. Information | |
| Section 14.5/Determination of Sample Size | regarding the analysis will be provided in the Statistical Analysis Plan. Subjects who participated in PAL-002 or PAL-004 may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy. | 1, 4 |
| Section 14.7/Interim Analyses | At least one interim analysis may be performed by the sponsor during the study. Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC). | 27 |
| Section 20/References | Lapis et al., Long-term correction of PKU in the Pahenu2 mouse by mutant and chemically modified forms of Phenylalanine Ammonium Lyase. The American Society of Human Genetics, 57th Annual Meeting, 2007 | 27 |



## CLINICAL STUDY PROTOCOL

Study Title: Long-term Extension of a Phase 2, Open-Label,

Dose-Finding Study to Evaluate the Safety, Efficacy, and

Tolerability of Multiple Subcutaneous Doses of

rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003

Investigational Product: rAvPAL-PEG (PEGylated recombinant Anabaena

variabilis phenylalanine ammonia lyase)

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria

Sponsor: BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Development Phase: Phase 2

Sponsor's Responsible

Medical Officer: , Clinical Sciences

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Duration: Up to 60 months or until study is terminated

Dose: 0.001 to a maximum weekly dose of 5.0 mg/kg

Date of Original Protocol:

October 08, 2008

Date of Amendment 1:

February 09, 2009

Date of Amendment 2:

October 30, 2009

May 04, 2011

Date of Amendment 4:

June 7, 2012


May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.



BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.

## CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

**Amendment: 4** 

**Date: June 7, 2012** 

## RATIONALE AND SUMMARY OF CHANGES

The protocol for Study PAL-003 is being amended to make the following changes:

1. Assessment of spot urine albumin/creatinine ratio has been added at study entry for newly enrolled subjects. In addition, all subjects will now have spot urine albumin/creatinine ratio assessed monthly after study entry. Complements (C3 and C4) will also be collected and assessed at study entry and every 3 months for all subjects; if complement levels are abnormal upon assessment, sampling will be performed monthly.

Rationale for change: The urine albumin/creatinine ratio and C3 and C4 tests have been added because they are measures of potential renal injury resulting from an immunologic reaction to rAvPAL-PEG. Several subjects currently being treated with rAvPAL-PEG have developed antibodies to rAvPAL-PEG and evidence of consumption of complement. While no subject in a rAvPAL-PEG study has had clinical laboratory evidence of renal injury as of May 2012, these tests have been added to increase detection of sensitivity to renal injury and to evaluate the potential for a clinically meaningful safety signal.

2. Subjects who meet the criteria for blood Phe levels and rAvPAL-PEG dose will now have their blood Phe concentration collected monthly rather than weekly.

Rationale for change: Subjects will have their blood Phe concentration assessed monthly versus weekly if they have been on a stable dose of rAvPAL-PEG (ie, no dose change in the last 2 weeks) and have had a phenylalanine (Phe) level at or below target range (60-600  $\mu$ mol/L) for 2 consecutive weeks, which is evidence that the dose-adjustment period has ended. For such subjects, assessment of blood Phe performed monthly is sufficient. However, if a subject's blood Phe increases to >600  $\mu$ mol/L or decreases to  $\leq$ 30  $\mu$ mol/L for any of the monthly blood Phe draws, that subject should perform weekly blood Phe draws until the rAvPAL-PEG dose has been adjusted and the Phe level returns to within the protocol-defined target range for at least 2 weeks.

|----------|------------|--------|

3. Information regarding hypersensitivity reactions and rAvPAL-PEG treatment, including how to treat hypersensitivity reactions, has been updated.

Rationale for change: As of May 2012, a total of 70 subjects have been administered rAvPAL-PEG in the Phase 1 (PAL-001) and Phase 2 (PAL-002 and -004) studies, including this extension study. With the information from these 70 subjects, there is a better understanding of the hypersensitivity reactions and rAvPAL-PEG treatment. Information regarding treatment with rAvPAL-PEG and subject care following a hypersensitivity reaction has been modified based on this additional information.

4. A fixed dose of rAvPAL-PEG will be administered in this study. Additionally, a higher concentration of rAvPAL-PEG (15 mg/ml vs. 10 mg/ml) will be administered. Subjects who have demonstrated efficacy (ie, Phe within target range 60-600 μmol/L) for at least two consecutive Phe assessments may convert their weight-based rAvPAL-PEG dose to a fixed dose and may also divide their weekly dose into a 7-days-a-week dosing regimen.

Rationale for change: The Phase 3 rAvPAL-PEG program will be conducted using a rAvPAL-PEG dosing concentration of 15 mg/ml, a fixed dose, and a 7-days-a-week dosing regimen. This extension study is being amended to incorporate the planned Phase 3 dosing regimen and concentration. Fixed dosing will simplify the dosing regimen to enable greater convenience for administration amongst the PKU patient population, especially for patients with significant neurocognitive dysfunction. The fixed doses proposed in this study are based on an average subject weight of 80 kg (based on the subjects in previous rAvPAL-PEG studies). Efficacy information regarding the fixed doses will be collected in this study and the Phase 2 study, 165-205. Subjects who are on a fixed-dose regimen will be monitored for safety per the safety plan outlined in the protocol. The 15 mg/ml rAvPAL-PEG formulation is more concentrated than the 10 mg/ml formulation, allowing for fewer injections per dose. It is hypothesized that hypersensitivity reactions could be related to maximum plasma concentration (C<sub>max</sub>); therefore, subjects who qualify for home or self administration may divide their weekly dose for administration up to 7 days per week.

5. A pharmacokinetics (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. A corresponding PK substudy objective has been added.

Rationale for change: Subjects who are being treated with an efficacious dose of rAvPAL-PEG (ie, have received the same rAvPAL-PEG dose for at least 2 consecutive weeks) and for whom no further dose modifications are planned will qualify for the PK substudy. 

|----------|------------|--------|

Single-dose PK data have been collected from the Phase 1 study, PAL-001; however, there is little multiple-dose PK data when a stable dosing regimen has been implemented. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved and maintained Phe reduction to within the protocol-defined target range.

6. The previous PK substudy that required stopping and restarting rAvPAL-PEG dosing has been removed. No subjects were enrolled into this PK substudy.

Rationale for change: The previous PK substudy was designed to examine the effect of rAvPAL-PEG dosing interruptions on safety, efficacy, PK, and immune response. This substudy has been discontinued because it requires subjects to discontinue treatment with rAvPAL-PEG, which would halt any Phe reduction benefits that may have occurred with treatment. The corresponding substudy objectives have been removed. Unscheduled dose interruptions may still occur due to adverse events per the Investigator and the Sponsor's Medical Officer.

7. Finger stick Phe assessments have been removed.

Rationale for change: The plasma Phe samples currently implemented in the study provide sufficient assessment of blood Phe levels without subjecting subjects to the additional and painful finger stick procedure. The site staff may perform assessments of Phe levels at the local laboratory if needed.

- 8. Guidance for treating subjects who develop hypophenylalaninemia has been added. Rationale for change: Although there is no evidence in the literature that low Phe is of clinical significance in adults, it is hypothesized that sustained low blood Phe is a clinical concern because Phe is an essential amino acid. Guidelines for treating subjects whose serum Phe levels reach  $\leq 30~\mu mol/L$  for a minimum of 1 month have now been included in the study.
- 9. A blood draw has been removed for subjects who enroll into PAL-003 from a previous rAvPAL-PEG study. Subjects who have performed a blood draw upon completion of a previous rAvPAL-PEG study do not need to perform another blood draw at the Screening Visit of this study if the blood draw was performed within 28 days. Safety and efficacy information are not expected to change in the 28 days from completion of a previous rAvPAL-PEG study and the start of this study.

Rationale for change: Currently, subjects in Studies PAL-002 and PAL-004 immediately enroll into the PAL-003 extension study (ie, do not stop rAvPAL-PEG dosing). The PAL-003 protocol required a blood draw to be performed as part of screening that was

|----------|------------|--------|

similar to the end-of-study blood draw performed for Studies PAL-002 and PAL-004. When subjects enroll over into Study PAL-003 within 28 days of completing a previous rAvPAL-PEG study, the screening blood draw is not needed. Safety and efficacy information is not expected to change in the 28 days from completion of a previous rAvPAL-PEG study and the start of this study.

- 10. Information regarding the management of allergic reactions has been updated. Rationale for change: Administration of oral or IV glucocorticoids has been added as a recommended treatment.
- 11. The inclusion criteria have been modified to allow enrollment of subjects from a Phase 2 rAvPAL-PEG study.

Rationale for change: This change will allow enrollment of subjects who complete Study 165-205.

12. Assessment of urinalysis test results has been moved from the local laboratory to the central laboratory.

Rationale for change: This change will help standardize test results across sites.

13. Subject weight will now be measured monthly rather than weekly.

Rationale for change: Because the study is moving from weight-based dosing to a fixed dosing regimen (see amendment item #5 above), there is no need to obtain weight on a weekly basis.

14. Subject diet diaries will be assessed monthly rather than weekly.

Rationale for change: Weekly diet diary assessment provides no added benefit to safety or efficacy when compared with monthly diet diaries. Monthly diet diary assessments will provide sufficient safety and efficacy information while increasing feasibility of completion for sites and subjects.

15. Information regarding clinical rAvPAL-PEG studies has been updated.

Rationale for change: Information regarding Studies PAL-002 and -004 have been updated, and information regarding Study 165-205 has been added.

16. Administrative revisions have been made to improve clarity and consistency. Specific revisions to the text of each section of the protocol (since the protocol amendment finalized on 4 May 2011), including the Synopsis, are outlined in Section 24.
|-------------------|
|-------------------|

### 2 SYNOPSIS

| NAME OF COMPANY BioMarin Pharmaceutical Inc. | SUMMARY TABLE Referring to Part of the | FOR NATIONAL<br>AUTHORITY USE |
|---|---|---|
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


**STUDY SITES**: Approximately 20 centers in the United States

PHASE OF DEVELOPMENT: Phase 2

### **STUDY RATIONALE:**

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205. Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for

|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

## **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

### STUDY DESIGN AND PLAN:

This is a long-term extension of rAvPAL-PEG Phase 2 studies in approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 5.0 mg/kg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either

| BIOMARIN <sup>®</sup> PAL-003 A4 Page 8 |
|-----------------------------------------|
|-----------------------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 µmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks). Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per

| BEOMARIN <sup>®</sup> PAL-003 A4 | Page 9 |
|----------------------------------|--------|
|----------------------------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

- A subject will continue in PAL-003 until one of the following occurs:
- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator.
- The subject has completed the study through the Month 60 visit.
- The study is terminated.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

## PAL-003 Substudy

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed.

### **Dose Modifications:**

### Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Sponsor's Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

• The dose may be increased by increments of no more than 10-fold higher than the subject's

|-----------------------------|
|-----------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

current dose.

- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg)) or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject.
- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg. Subjects who increase their dose frequency will have additional assessments performed (Interim Dosing Visit).
- When a dose is increased, the subject must be observed for 30-60 minutes following the first
  modified dose administration. Subjects who increase their dose frequency do not need to be
  observed following injection of study drug if the increase in frequency does not increase the
  overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

### Dose Decrease Methodology

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for safety (ie, any adverse event that may be improved with a lower, more frequent dose).

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L as measured by serum Phe levels for a minimum of 1 month), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for

| BIOMARIN <sup>®</sup> PAL-003 A4 Page 11 |
|------------------------------------------|
|------------------------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

PKU disease management, subject diet should be monitored by a dietician).

### **Safety Assessment Criteria:**

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Sponsor's Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level.

### **Stopping Criteria:**

If 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will be evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate.

### NUMBER OF SUBJECTS PLANNED:

Approximately 100 subjects.

## DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.

|--------------------|
|--------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.

|----------|------------|---------|
|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from a previous rAvPAL-PEG study.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

## INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing  $1.5 \pm 0.2$  mL to deliver either 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration) or 15 mg or rAvPAL-PEG per 1 mL (15 mg/mL protein concentration). Each vial is filled with  $1.5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies will be dosed with the same or higher dose than the dose that was administered upon completion of that study provided that there was no interruption in dosing. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Sponsor's Medical Officer, based upon the subject's response to doses.

### **Fixed Dosing**

Subjects who have demonstrated efficacy (ie, blood Phe within the target range of  $60\text{-}600~\mu\text{mol/L}$  for at least 2 consecutive weeks) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects should convert their weight-based dose using the following table:

|----------|------------|---------|
|----------|------------|---------|

NAME OF COMPANY **SUMMARY TABLE** FOR NATIONAL BioMarin Pharmaceutical Inc. Referring to Part of the **AUTHORITY USE** Dossier: 105 Digital Drive **ONLY:** Novato, CA 94949 Volume: NAME OF FINISHED PRODUCT: Page: rAvPAL-PEG (PEGylated recombinant Reference: Anabaena variabilis phenylalanine ammonia lyase) NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase

| Weight-based dose<br>(mg/kg) | Equivalent fixed dose (mg) | Vol for 10 mg/ml<br>concentration (ml) | Vol for 15 mg/ml<br>concentration (ml) |
|---|---|---|---|
| 0.03 | 2.5 | 0.25 | 0.17 |
| 0.06 | 5 | 0.5 | 0.33 |
| 0.12 | 10 | 1 | 0.67 |
| 0.25 | 20 | 2 | 1.33 |
| 0.5 | 40 | 4 | 2.67 |
| 1.0 | 75 | 7.5 | 5 |
| 2.0 | 150 | 15 | 10 |
| 3.0 | 225 | 22.5 | 15 |
| 4.0 | 300 | 30 | 20 |
| 5.0 | 375 | 37.5 | 25 |

## **DURATION OF TREATMENT:**

Up to 60 months.

## REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

## **CRITERIA FOR EVALUATION:**

### **Efficacy**:

Blood Phe concentrations will be measured.

### **Immunogenicity**:

The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-PEG neutralizing antibodies, and anti-PEG-PAL IgE) will be assessed.

## Safety:

|--|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. | SUMMARY TABLE Referring to Post of the | FOR NATIONAL |
|---|---|---|
| | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs, ECG results, X-ray results, and laboratory test results.

### Pharmacokinetic:

Plasma concentrations of rAvPAL-PEG will be measured for subjects participating in the Substudy.

#### STATISTICAL METHODS:

## Sample Size:

Subjects who participated in a previous rAvPAL-PEG study may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

### **Safety Analysis:**

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by—subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, ECG results, and X-ray results will also be provided.

### **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be

|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 60-600 µmol/L will be summarized by each scheduled time point.

## **Exploratory Analysis**:

For subjects who have received any study drug in this study with any post-treatment blood Phe concentration measurements and diet diary information, the relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will be explored.

### **Substudy Analysis**:

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

### Pharmacokinetic Analysis:

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F).




# 3 TABLE OF CONTENTS

| 1 | TIT | LE PAG | E | 1 |
|---|---|---|---|---|
| 2 | SYN | NOPSIS. | | <i>6</i> |
| 3 | TAI | BLE OF | CONTENTS | 17 |
| 4 | LIS | T OF AF | BBREVIATIONS AND DEFINITIONS OF TERMS | 21 |
| 5 | ETF | HCS | | 25 |
| | 5.1 | Institut | tional Review Board or Ethics Committee | 25 |
| | 5.2 | Ethical | Conduct of Study | 25 |
| | 5.3 | Subjec | t Information and Informed Consent | 26 |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 27 |
| 7 | INT | RODUC | CTION | 28 |
| | 7.1 | Noncli | nical Studies | 28 |
| | 7.2 | Previo | us Clinical Studies | 30 |
| | | 7.2.1 | Phase 1 Study PAL-001 | 30 |
| | | 7.2.2 | Phase 2 Studies PAL-002, PAL-004, and 165-205 | 31 |
| | 7.3 | Study 1 | Rationale | 32 |
| | 7.4 | Summa | ary of Overall Risks and Benefits | 34 |
| | | 7.4.1 | Toxicity Due to Exposure to PEG | 34 |
| | | 7.4.2 | Toxicity Due to an Immunologic Reaction | 34 |
| 8 | STU | JDY OB | JECTIVES | 39 |
| 9 | INV | ESTIGA | ATIONAL PLAN | 40 |
| | 9.1 | Overal | l Study Design and Plan | 40 |
| | | 9.1.1 | Management of Local and Systemic Reactions to rAvPAL-PEG | 48 |
| | | 9.1.2 | Dose Modifications | 53 |
| | | 9.1.3 | Safety Assessment Criteria | 55 |
| | | 9.1.4 | Stopping Criteria | 55 |
| | 9.2 | | sion of Study Design, Including Choice of Control Group | |
| | 9.3 | Selecti | on of Study Population | 55 |

| BIOM | 1AR | N |
|------|-----|---|
|------|-----|---|


| | | 9.3.1 | Inclusion Criteria | 55 |
|---|---|---|---|---|
| | | 9.3.2 | Exclusion Criteria | 56 |
| | | 9.3.3 | Removal of Subjects from Treatment or Assessment | 57 |
| | | 9.3.4 | Subject Identification and Replacement of Subjects | 58 |
| | 9.4 | Treatme | ents | 58 |
| | | 9.4.1 | Treatments Administered | 60 |
| | | 9.4.2 | Identity of Investigational Product (IP) | 60 |
| | | 9.4.3 | Storage | 61 |
| | | 9.4.4 | Directions for Administration | 61 |
| | | 9.4.5 | Method of Assigning Subjects to Treatment Groups | 63 |
| | | 9.4.6 | Selection of Doses Used in the Study | 64 |
| | | 9.4.7 | Blinding | 64 |
| | | 9.4.8 | Prior and Concomitant Medications | 64 |
| | | 9.4.9 | Treatment Compliance | 65 |
| | | 9.4.10 | Dose Interruption and Missed Doses | 65 |
| | 9.5 | Investig | gational Product Accountability | 65 |
| | | 9.5.1 | Return and Disposition of Clinical Supplies | 66 |
| | 9.6 | Dietary | or Other Protocol Restrictions | 66 |
| | 9.7 | Efficacy | y and Safety Variables | 67 |
| | | 9.7.1 | Efficacy and Safety Measurements Assessed | 67 |
| | | 9.7.2 | Efficacy Variable | 68 |
| | | 9.7.3 | Pharmacokinetic Variables | 69 |
| | | 9.7.4 | Exploratory Efficacy Variable | 69 |
| | | 9.7.5 | Safety Variables | 69 |
| | | 9.7.6 | Clinical Laboratory Assessments | 70 |
| 10 | REP | ORTING | G ADVERSE EVENTS | 73 |
| | 10.1 | Adverse | e Events | 73 |
| | 10.2 | Serious | Adverse Events | 76 |
| | 10.3 | Dramar | nev | 77 |

| BIOM | 1AR | IN |
|------|-----|----|
|------|-----|----|


| | 10.4 Urgent Safety Measures | 77 |
|----|------------------------------------------------------|----|
| | 10.5 BioMarin Pharmacovigilance Contact Information | 78 |
| 11 | APPROPRIATENESS OF MEASUREMENTS | 79 |
| | 11.1 Safety and Pharmacokinetics | 79 |
| | 11.2 Diet Diary | 79 |
| 12 | STUDY PROCEDURES | 80 |
| | 12.1 Prestudy | 80 |
| | 12.2 Screening Visit | 80 |
| | 12.3 Treatment Period | 80 |
| | 12.3.1 Day 1 (Week 1) | 81 |
| | 12.3.2 Weekly Visits | 81 |
| | 12.3.3 Substudy Visits | 82 |
| | 12.3.4 Monthly Visits (Week 4, 8, 12, etc) | 82 |
| | 12.3.5 Quarterly Visits (Week 12, 24, 36, etc) | 83 |
| | 12.3.6 Interim Dosing Visit | 83 |
| | 12.3.7 Weekly Telephone Visit | 84 |
| | 12.3.8 Unscheduled Hypersensitivity Reaction Visit | 84 |
| | 12.4 Early Termination Visit | 85 |
| | 12.5 Final Follow-up Visit | 86 |
| 13 | DATA QUALITY ASSURANCE | 87 |
| 14 | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 88 |
| | 14.1 Statistical and Analytical Plans | 88 |
| | 14.2 Safety Analysis | 88 |
| | 14.3 Pharmacokinetic Analysis | 88 |
| | 14.3.1 Pharmacokinetic Substudy Analysis | 89 |
| | 14.4 Efficacy Analysis | 89 |
| | 14.5 Determination of Sample Size | 89 |
| | 14.6 Handling of Missing Data | 89 |
| | 14.7 Interim Analyses | 89 |

|--|----------|------------|---------|
|--|----------|------------|---------|

| | 14.8 Changes in the Conduct of the Study or Planned Analyses | 90 |
|---|---|---|
| 15 | DATA MONITORING COMMITTEE (DMC) | 91 |
| 16 | COMPENSATION, INSURANCE, AND INDEMNITY | 92 |
| 17 | CASE REPORT FORMS AND SOURCE DOCUMENTS | 93 |
| 18 | STUDY MONITORING AND AUDITING | 95 |
| 19 | RETENTION OF RECORDS | 96 |
| 20 | USE OF INFORMATION AND PUBLICATION | 97 |
| 21 | REFERENCES | 98 |
| 22 | INVESTIGATOR RESPONSIBILITIES | 100 |
| | 22.1 Conduct of Study and Protection of Human Subjects | 100 |
| 24 | PROTOCOL AMENDMENT TEXT REVISIONS | 102 |
| LIS | ST OF TABLES | |
| Tal | ble 9.1.1: Schedule of Events | 42 |
| Tal | ble 9.1.2: PK Substudy Dosing Regimens | 47 |
| Tal | ole 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen | 62 |
| Tal | ble 9.4.4.2: Number of Injections Required For an Individual Weighing 80 kg | 63 |
| Tal | ble 9.7.1.1: Summary of Laboratory Assessments | 67 |
| Tal | ble 9.7.6.1: Clinical Laboratory Tests | 71 |

# LIST OF FIGURES




### 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

## <u>Abbreviations</u>

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase

AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

 $AUC_{0-7 \, days}$  area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen

°C degree Celsius

C<sub>3</sub> complement 3

C<sub>4</sub> complement 4

CBC complete blood count

CD Compact disk

CFR Code of Federal Regulations

CH50 total hemolytic complement

C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form

CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

|----------|------------|---------|

DBP diastolic blood pressure

DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up

g gram

GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure

ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IgE immunoglobulin E

IgG immunoglobulin G

IgM immunoglobulin M

IP investigational product

IRB Institutional Review Board

IV intravenous

kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

|----------|------------|---------|

NAb neutralizing antibodies

NCI National Cancer Institute

NOAEL no observable adverse effect level

OTC over the counter

PAH phenylalanine hydroxylase

PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator

PK pharmacokinetics

PKU phenylketonuria

rAvPAL-PEG recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG

RBC red blood cell

SAE serious adverse event

SAP Statistical Analysis Plan

SBP systolic blood pressure

SC subcutaneous

SD standard deviation

SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase

SGPT serum glutamic pyruvate transaminase

US United States

WBC white blood cell

| PAL-003 A4 Page 24 | BIOMARIN | PAL-003 A4 | Page 24 |
|--------------------|----------|------------|---------|
|--------------------|----------|------------|---------|

Definition of Terms:

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.

|--------------------|
|--------------------|

### 5 ETHICS

### 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

## 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will 

|--|

provide written, informed consent before any study-related tests or evaluations are performed.

## 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR Part 50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



### 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Regulatory Affairs Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations and urinalysis. Pharmacokinetic (PK) analysis will be performed by BioMarin.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.

|----------|------------|---------|--|

### 7 INTRODUCTION

A comprehensive review of PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

### 7.1 Nonclinical Studies

The nonclinical program for rAvPAL-PEG has characterized the pharmacology, pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC route of administration. Pharmacology was assessed in the BTBR *Pah*<sup>enu2</sup> (ENU2) mouse model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to 2000 μM) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to male ENU2 mice, plasma Phe concentrations decreased from approximately 2000 μM to < 200 μM after 2 dose administrations. An attenuated reduction of blood Phe was seen between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe < 200 μM over the entire week, which continued for a total of 15 weeks.

In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a 2-4 week dose interruption and an 11-week dose interruption. Following both dose interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A similar interim attenuated response was observed with the longer dose interruption of approximately 11 weeks. In both of these assessments, no safety issues were noted upon re-starting dosing with rAvPAL-PEG (Lapis, 2007, ASHG 57th Annual Meeting).

Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No respiratory or central nervous system (CNS) effects were seen with SC administration of rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV effects of rAvPAL-PEG administered subcutaneously.

Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats and cynomolgus monkeys. The elimination half-life  $(t_{1/2})$  values of rAvPAL-PEG administered to 

|--------------------|
|--------------------|

normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and 44 hours, respectively, and exhibited modest area under the plasma concentration-time curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the  $t_{1/2}$  was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum observed plasma concentration ( $C_{max}$ ), along with a long  $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) the AUC and the  $C_{max}$  are roughly linearly proportional.

Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given ≥ 3 mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey.



### 7.2 Previous Clinical Studies

The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002, Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience as of JAN2011 from this ongoing study and the other ongoing Phase 2 studies, PAL-002 and PAL-004.

## **7.2.1 Phase 1 Study PAL-001**

The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations.

The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 µmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG.

Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows:

- rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg.
- For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level for these 5 subjects was 1113 µmol/L.
- Overall, no clinically significant reductions in blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, 0.01, and 0.03 mg/kg.

|--------------------|
|--------------------|

• For subjects who were administered rAvPAL-PEG at the 3 higher dose levels (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration levels, the calculated PK parameters were a mean T<sub>max</sub> of 89-106 hours, a t<sub>1/2</sub> of 46-120 hours, and an AUC<sub>0-t</sub>, and C<sub>max</sub> that were proportional with dose. Drug exposure was slightly increased with increased dose.

## 7.2.2 Phase 2 Studies PAL-002, PAL-004, and 165-205

Currently, rAvPAL-PEG is being investigated in three Phase 2 clinical trials (PAL-002 and PAL-004). As of May 2012, a total of 70 subjects have been administered rAvPAL-PEG in a rAvPAL-PEG Phase 2 study.

In PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU), approximately 55 subjects will be enrolled and will be administered multiple doses of rAvPAL-PEG up to 5.0 mg/kg/week. PAL-002 is a 2-part study. In Part 1, subjects will be assigned to 1 of 4 rAvPAL-PEG dose cohorts (0.001, 0.003, 0.01, 0.1 mg/kg, or 1.0 mg/kg). rAvPAL-PEG will be administered at a fixed weekly dose of 0.001 mg/kg (Cohort 1), 0.003 mg/kg (Cohort 2), 0.01 mg/kg (Cohort 3), 1.0 mg/kg (Cohort 4), or 0.1 mg/kg (Part 1 Substudy) for 8 weeks. In Part 2, all subjects who complete Part 1 will be administered an adjustable dose of rAvPAL-PEG for up to an additional 8 weeks. The dose administered in Part 2 may be adjusted by dose level and/or dose frequency to reach a target blood Phe concentration of 60-600 μmol/L.

Study PAL-003 (Long-Term Extension of a Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU) is an extension study of PAL-002, PAL-004 and 165-205 (A Phase 2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate Safety, Efficacy and Tolerability of Subcutaneously Administered rAvPAL-PEG in Patients with PKU for 24 Weeks). Once subjects have completed a previous rAvPAL-PEG study, they have the option to enroll into PAL-003 and to continue to receive doses of rAvPAL-PEG for up to an additional 60 months.

Study PAL-002 was initiated in September 2009 and is ongoing. The primary objective of this study is to evaluate the effect of multiple doses of rAvPAL-PEG on blood Phe concentrations in subjects with PKU for up to 16 weeks of treatment. The secondary objectives of the study are (1) to evaluate the safety and tolerability of SC injections of multiple dose levels of rAvPAL-PEG, (2) to evaluate the antibody response to rAvPAL-PEG,

|--------------------|
|--------------------|

and (3) to evaluate the PK profile of rAvPAL-PEG in subjects with PKU. The study protocol was amended (30APR2010) to include a substudy of an additional rAvPAL-PEG dose level (0.1 mg/kg/week) that reduced blood Phe concentrations to clinically significant levels in the Phase 1 study, PAL-001. The protocol was amended again (28MAR2011) to increase the starting dose for Cohort 4 from 0.03 mg/kg/week to 1.0 mg/kg/week. As of JAN2011, 33 subjects have been enrolled into the study and all 10 subjects of the substudy have been dosed with 0.1 mg/kg rAvPAL-PEG. Additional information about the safety reported as of JAN2011 is provided in Section 7.4.2.

Study PAL-004 is designed to determine if daily administration of rAvPAL-PEG at daily dose levels (0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day) is safe and effective in reducing and maintaining consistent blood Phe concentrations in subjects with PKU. It is hypothesized that a higher starting dose and frequency will reduce blood Phe concentrations to near-normal levels in a timely manner and will provide the greatest clinical benefit. Considering the concentration and volume of drug that is administered subcutaneously, the only way to increase the rAvPAL-PEG dose is via daily administration. Therefore, in Study PAL-004, a higher starting dose of 0.4 mg/kg will be administered 5 days a week (referred to as daily), a dosing regimen that has been observed to be tolerated and to reduce blood Phe concentrations to clinically meaningful levels in previously exposed subjects in this study. Following completion of Study PAL-004, subjects have the option to enroll into this study and to continue to receive doses of rAvPAL-PEG for up to an additional 60 months.

Study 165-205 is a Phase 2 study using a subject-driven dose modification schema to assess safety. In addition, fixed dosing at a drug concentration of 15 mg/mL rAvPAL-PEG will be assessed. As of May 2012, enrollment of subjects is underway for this study.

In this study, subjects who completed a previous rAvPAL-PEG study will continue to be administered the same rAvPAL-PEG dose that was administered in the previous study. If the safety, PK, and blood Phe concentration results from the previous study indicate that the appropriate level of PEGylation and dosing regimen differs from that administered in the previous study, the PEGylation and/or dosing regimen administered in this study may change.

### 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH. Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally 

|--|

elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan<sup>®</sup> is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. rAvPAL-PEG is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is

|--|

little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

This study is an extension of previous rAvPAL-PEG studies. Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

# 7.4 Summary of Overall Risks and Benefits

It is not expected that data from previous rAvPAL-PEG studies will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

## 7.4.1 Toxicity Due to Exposure to PEG

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg rAvPAL-PEG SC. In rats, both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1).

In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

## 7.4.2 Toxicity Due to an Immunologic Reaction

The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). In vivo 

|--------------------|
|--------------------|

and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylation does not eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing the immunogenicity of the molecule, it is reasonable to expect that some individuals may exhibit immune responses upon exposure to the drug. These immune responses may be clinically irrelevant, cause symptoms of various degrees, or lead to neutralization of biological activity. Subjects participating in clinical trials will be monitored closely with specific antibody titers, sedimentation rates, and complete blood counts (CBCs).

As of May 2012, a total of 70 subjects have been administered rAvPAL-PEG in the single-dose, Phase 1 study (PAL-001) and in the repeat -dosing Phase 2 studies (PAL-002, PAL-004, and PAL-003). The dose levels in the repeat-dosing studies range from 0.001 to 5.0 mg/kg/week administered in various frequencies (including 5 days a week). The most clinically significant AEs have been hypersensitivity reactions that have led to dosing interruptions and reductions. Most of the hypersensitivity reactions have been nonserious and mild-to-moderate in severity.

A total of 4 SAEs have been reported in the previous rAvPAL-PEG studies. Of these 4 SAEs, 3 have been reported as related to rAvPAL-PEG. Two of the study-drug related SAEs occurred in Study PAL-001. Both of these SAEs occurred in subjects in the lower dose cohorts: an SAE of hypersensitivity reaction in a subject in the 0.001 mg/kg cohort and an SAE of anaphylactic reaction (urticaria) in a subject in the 0.01 mg/kg cohort. Neither SAE was severe or resulted in discontinuation from the study, and both of the SAEs resolved. There were no SAEs in subjects in the higher dose cohorts (0.03 mg/kg and 0.1mg/kg) in PAL-001. The third study drug-related SAE (angioedema) occurred in a subject in Study PAL-004. The fourth SAE (urticaria, dehydration) was reported as not related to study drug and occurred in a subject in Study PAL-002. There have been no reports of anaphylaxis for any subject treated with rAvPEG-PAL (as of January 2012).

Subjects who have a systemic clinical reaction at any time during this study may undergo a series of assessments to monitor safety, including assessment of complements, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and IgE antibodies. Reintroduction of rAvPAL-PEG dosing after a reaction will depend on clinical assessments and available laboratory data, such as chemistry and urine studies, to ensure that there has been no

|--------------------|
|--------------------|

end-organ damage prior to resuming treatment with rAvPAL-PEG. As of May 2012, antibody titers, including positive IgE titers, have not been predictive of future clinical reactions when dosing with rAvPAL-PEG. Additionally, subjects will be premedicated to prevent or mitigate risk of hypersensitivity reactions (refer to Section 9.1.1.3.3).

PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.), (Harris, 2003, Nat.Rev.Drug Discov.), however, antibodies against PEG may form when PEG is bound to compounds. (Harris, 2003, Nat.Rev.Drug Discov.), (Richter, 1983, Int.Arch.Allergy Appl.Immunol.). In some instances, development of such antibodies did not result in any significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.). Administration of rAvPAL-PEG may lead to anti-PEG antibody formation, and the duration of this possible effect is not known. Subjects in the Phase 2 rAvPAL-PEG studies have developed both anti-PEG IgM and anti-PEG IgG antibodies. Antibody formation\_may limit a subject's future ability to be treated with other PEG-containing (eg, Depo-Provera) or PEGylated (eg, PEG-interferon) injectable drugs. It is therefore recommended that any PEG-containing injectable drug administered to subjects after completion of this study be done under medical observation.

## 7.4.2.1 Systemic Skin Reactions

Two out of 25 subjects who were enrolled in Study PAL-001 and received the protocol-defined single dose of rAvPAL-PEG reported systemic skin reactions (generalized skin rash) that were attributed to treatment with study drug. One subject received a single dose of 0.001 mg/kg rAvPAL-PEG, and the other subject received a single dose of 0.01 mg/kg rAvPAL-PEG. One of these events was reported as serious, and the other was reported as nonserious; both events were reported following administration of Depo-Provera injections (medroxyprogesterone injection), an injectable contraception. These allergic reactions are thought to be related to the PEG molecules that are found in both the study drug, rAvPAL-PEG, and Depo-Provera. These reactions are not likely to be experienced concurrent with other birth control medications.

The 2 subjects were administered study drug during PAL-001 and then experienced an allergic reaction following an injection of Depo-Provera. The symptoms of the reactions were hives on the arms and legs and difficulty breathing. The symptoms for both subjects

|--------------------|
|--------------------|

Both subjects were examined by an allergy specialist after they completed participation in PAL-001. A skin prick test with Depo-Provera was administered as part of this examination. One subject had a mild allergic reaction to the test; however, no further reactions or complications were reported following subsequent administration of a full dose of Depo-Provera. Upon study completion, the subject continued to receive regular doses (every 3 months) of Depo-Provera, and no further reactions were reported. The second subject also had a positive reaction to Depo-Provera following administration of the skin prick test. When a subsequent full dose of Depo-Provera was administered, developed hives, itching, and chills. The subject's symptoms resolved within 1 day of taking medication prescribed by an allergist. See Section 7.2.1 for the results from Study PAL-001.

The active drug substance in rAvPAL-PEG is a bacterial protein that may elicit immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and others. The results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys indicated the formation of anti-rAvPAL antibody titers that did not correspond with observations of injection-site reactions. Quantitation of anti-PEG titers were not assessed in the chronic repeat-dose studies in the rat and monkey. Although results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys did not indicate signs of immune-mediated toxicities, it is possible that the physio-chemical properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG in humans. It is currently unknown whether administration of PEG-containing drugs, such as Depo-Provera, has a sensitizing effect to PEG in rAvPAL-PEG when administered in humans. Because the exact basis for these reported events and their duration is not known, the use of PEG-containing injectable drugs prior to, during, and after this study is prohibited as a precautionary measure (refer to Section 9.3.2 and Section 9.4.8).

# 7.4.2.2 Management of Allergic Reactions

Allergic reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 30-60 minutes post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of allergic reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the

rAvPAL-PEG injection. Subjects who qualify for self administration of study drug will be provided with emergency resuscitation instructions (refer to Section 9.4 and the Subject Self-Administration Training Materials).

In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for immunology studies and complement testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of allergic symptoms:

- Maintain the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oral or IV glucocorticoids.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment (eg, acetaminiophen or ibuprofen).
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. An allergy and/or immunology consultation should be sought if necessary. Information regarding the management of local skin, large local skin, and systemic reactions is provided in Section 9.1.1. Detailed instructions for the management of allergic reactions are provided in the Study Reference Manual.



### 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objective is as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

|----------|------------|---------|

### 9 INVESTIGATIONAL PLAN

## 9.1 Overall Study Design and Plan

This is a long-term extension of rAvPAL-PEG Phase 2 studies in approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 5.0 mg/kg/week), provided no dose-limiting toxicity was observed in a previous rAvPAL-PEG studies.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to clinic monthly for review with the clinical study staff.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self administration. Additional information is provided in the Subject Self-Administration Training Materials.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

| BIOMARIN PAL-003 A4 Page 41 | BIOMARIN <sup>®</sup> | PAL-003 A4 | Page 41 |
|-----------------------------|-----------------------|------------|---------|
|-----------------------------|-----------------------|------------|---------|

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 μmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 μmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks; refer to Section 9.4.4). Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 9.1.1 and Table 9.1.2. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator.
- The subject has completed the study through the Month 60 visit.
- The study is terminated.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed (refer to Table 9.1.2.

The Schedule of Events and PK substudy collection schedules are presented below in Table 9.1.1 and Table 9.1.2



**Table 9.1.1: Schedule of Events** 

| | | | Tr | eatment Per | riod <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly <sup>b</sup> | Monthly<br>(eg, Wk 4,<br>8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Interim<br>Clinician<br>Visit<br>(HHRN or<br>Site) | Final F/U<br>Visit | Self<br>Administra-<br>tion | Early<br>Term.<br>Visit | |
| Assessments and Events | Screening <sup>a</sup> | <b>D</b> 1 | Starting at Week 2 | Every 4th<br>week;<br>Perform<br>in<br>addition<br>to weekly<br>procedure<br>s | Every 12th week. Perform in addition to monthly procedures | | 1 week<br>after final<br>dose | | 4 weeks<br>after final<br>dose | Unsched.<br>Hyper.<br>Reaction<br>Visit. <sup>d</sup><br>Perform<br>within<br>48 hours |
| Informed consent | X | | | | | | | | | |
| Medical history, including allergy history, and demographics | X | | | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | | X | | X | | X | |
| Vital signs <sup>e</sup> | X | X | X | | | X | | | X | X |
| Weight | X | | | X | | | | | | |
| 12-lead ECG | X | | | | | | X | | X | |




| | | | Tr | eatment Per | riod <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | <b>Weekly</b> <sup>b</sup> | Monthly<br>(eg, Wk 4,<br>8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Interim<br>Clinician<br>Visit<br>(HHRN or<br>Site) | Final F/U<br>Visit | Self<br>Administra-<br>tion | Early<br>Term.<br>Visit | |
| Assessments and Events | Screening <sup>a</sup> | <b>D</b> 1 | Starting<br>at Week 2 | Every 4th<br>week;<br>Perform<br>in<br>addition<br>to weekly<br>procedure<br>s | Every 12th week. Perform in addition to monthly procedures | Up to daily | 1 week<br>after final<br>dose | | 4 weeks<br>after final<br>dose | Unsched. Hyper. Reaction Visit. <sup>d</sup> Perform within 48 hours |
| Clinical laboratory tests <sup>f</sup> | X | | | X | | | X | | X | $X^g$ |
| Complements C <sub>3</sub> and C <sub>4</sub> <sup>h</sup> | X | | | | X | | | | | X |
| Sedimentation rate | | X | | | X | | X | | X | X |
| Chest x-ray | X | | | X<br>(Week 48<br>visit only) | | | X | | X | |
| Urine pregnancy test <sup>i</sup> | X | X | | X | | | X | | X | |
| Injection-site inspectionj <sup>i j</sup> | | X<br>(postdose | X | | | X | X | X | X | X |




| | | | Tr | eatment Per | riod <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | <b>Weekly</b> <sup>b</sup> | 8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Interim<br>Clinician<br>Visit<br>(HHRN or<br>Site) | Final F/U<br>Visit | Self<br>Administra-<br>tion | Early<br>Term.<br>Visit | |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at Week 2 | Every 4th<br>week;<br>Perform<br>in<br>addition<br>to weekly<br>procedure<br>s | Every 12th week. Perform in addition to monthly procedures | Up to daily | 1 week<br>after final<br>dose | | 4 weeks<br>after final<br>dose | Unsched. Hyper. Reaction Visit. <sup>d</sup> Perform within 48 hours |
| Adverse events <sup>j, k</sup> | X | X | X | | 1 | X | X | X | X | X |
| Weekly phone call to self<br>admin participants only (to<br>assess AEs, Inj site reactions,<br>concomitant medications) | | | | | | | | X | X | |
| Concomitant medications <sup>j</sup> | X | X | X | | | X | X | X | X | X |
| Diet query | X | X | X | | | | X | | X | |
| 3-Day diet diary <sup>l</sup> | | | | X | | | X | | X | |
| Serum antibodies | | X | | X | | | X | | X | X |
| Plasma Phe and plasma | X | X | X | X <sup>m</sup> | | | X | | X | |




| | | | Tr | eatment Per | riod <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly <sup>b</sup> | Monthly<br>(eg, Wk 4,<br>8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Interim<br>Clinician<br>Visit<br>(HHRN or<br>Site) | Final F/U<br>Visit | Self<br>Administra-<br>tion | Early<br>Term.<br>Visit | |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at Week 2 | Every 4th week; Perform in addition to weekly procedure s | Every 12th<br>week.<br>Perform in<br>addition to<br>monthly<br>procedures | Up to daily | 1 week<br>after final<br>dose | | 4 weeks<br>after final<br>dose | Unsched. Hyper. Reaction Visit. <sup>d</sup> Perform within 48 hours |
| tyrosine <sup>m</sup> | | | | | | | | | | |
| Plasma PK sample | | X | Xº | | | | X | | X | X |
| Administer study drug <sup>n</sup> | | X | X | | | X | | X | | |
| Skin biopsy (optional; affected and not affected area) | | | | | | | | | | X |
| Serum tryptase level ° | | | | | | | | | | X |

AE, adverse event; C<sub>3</sub>, complement 3; C<sub>4</sub>, complement 4; CH50, total hemolytic complement; CRP, C-reactive protein; D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> A separate Screening visit for this study is required only if the time between completion of the previous rAvPAL-PEG study and enrollment into PAL-003 is greater than 28 days.




<sup>&</sup>lt;sup>b</sup> Weekly visits do not require an in-clinic visit if conducted by a home healthcare professional. Monthly visits must be performed in the clinic.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Refer to Section 9.1.1.3.3 and Section 12.3.8.

<sup>&</sup>lt;sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.

<sup>&</sup>lt;sup>f</sup> Clinical laboratory tests to include spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis. Urine microscopy will be performed if any urinalysis results are positive for hematuria. Refer to Table 9.7.6.1.

<sup>&</sup>lt;sup>g</sup> Subjects who have a systemic reaction or a large local reaction not contiguous with the injection site should be assessed for CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub> within 48 hours of the reaction.

<sup>&</sup>lt;sup>h</sup>Complement C<sub>3</sub> and C<sub>4</sub> will be collected at the Screening Visit and quarterly. Additional complement testing will be performed and as needed to resolve previous abnormal test results.

<sup>&</sup>lt;sup>i</sup> If positive or equivocal, perform serum pregnancy test.

<sup>&</sup>lt;sup>j</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm).

<sup>&</sup>lt;sup>j</sup> Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

<sup>&</sup>lt;sup>k</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug to the final study visit.

<sup>&</sup>lt;sup>1</sup> It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.

<sup>&</sup>lt;sup>m</sup> Samples should be drawn at least 2.5 hours after a meal. At the Investigator's discretion, blood Phe may be collected monthly rather than weekly, provided the subject satisfies the criteria in Section 9.7.2.1.

<sup>&</sup>lt;sup>n</sup> Dosing is up to 5.0 mg/kg/week, including subjects who receive more than 1 dose/week. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may be re-evaluated.

<sup>&</sup>lt;sup>o</sup> Mandatory for subjects who have a systemic reaction. Take sample immediately after reaction if possible.




**Table 9.1.2: PK Substudy Dosing Regimens** 

| Treatment Frequency | Plasma PK Sampling | Example |
|---|---|---|
| Subjects who are<br>administered study drug<br>once per week | Pre-dose and every 24 hours<br>thereafter (24, 48, 72, and 96 hours<br>when possible), and pre-dose of the<br>next weekly dose | If dosed on Monday: Obtain PK sample pre-dose when possible – pre-dose Monday, Tuesday, Wednesday, Thursday, Friday, and pre-dose the following Monday. No further PK substudy draws. |
| Subjects who are administered study drug two or three times per week | Pre-dose and every 24 hours during the longest period between doses, when possible, and pre-dose of the next dose. | If dosed on Monday, Thursday, and Friday: Obtain PK sample every 24 hours during the longest period between doses: Pre-dose Monday, Tuesday, Wednesday, and pre-dose Thursday. No further PK substudy draws. |
| Subjects who are administered study drug four to seven times per week. | Pre-dose and every 12 hours during the longest period between doses, when possible, then pre-dose of the next dose. | If dosed Monday through Friday: Obtain PK sample every 12 hours during the longest period between doses (Friday to Monday): pre-dose Friday, 12 hours post-dose Friday, Saturday (24 and 36 hours post dose), Sunday (48 and 60 hours post-dose), and pre-dose the following Monday. No further PK substudy draws. |



#### 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEG

Subjects who qualify for self administration of study drug will be provided with information and instruction with regard to management of local and systemic reactions (refer to the Subject Self-Administration Training Materials).

# 9.1.1.1 Subjects Who Have Had Previous Hypersensitivity Reactions to rAvPAL-PEG or a PEG-containing Product

Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from a previous rAvPAL-PEG study are excluded from participation in this study. Subjects who experienced a generalized skin rash are included in this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in a previous rAvPAL-PEG study are eligible to participate in this study. Subjects who have had a previous reaction and are deemed eligible for participation must be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing for the remainder of the study. The premedication dosage will be standard. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). Subjects may develop systemic, large local skin, or local skin reactions after enrollment in PAL-003. Refer to Section 9.1.1.2 for definitions of systemic and local skin reactions. For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1

# 9.1.1.2 Definition of Reaction and Hypersensitivity Reactions to rAvPAL-PEG Administered Subcutaneously

During Study PAL-003, subjects may experience hypersensitivity reactions to rAvPAL-PEG. The hypersensitivity reactions are defined as follows:

Local skin reaction:

• Skin signs or symptoms in 1 affected primary location, ie, hives, wheals, or swelling or an area of erythema, redness, induration, pain, or itching at or near the site of injection.

Large local skin reaction:



• Skin signs or symptoms, ie, hives, wheals, or swelling or an area of erythema, redness, or induration with pain or itching that extends beyond the site of injection by approximately 6 inches (15 cm) and/or signs or symptoms that are not contiguous to the injection site. These may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure and, therefore, will be managed as a systemic reaction when not contiguous to the injection site.

Systemic reaction (including generalized skin symptoms):

• Skin and non-skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological; and/or a fever attributed to treatment with rAvPAL-PEG ( ≥ 100.4°F or ≥ 38°C).

For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1



| BIOMARIN | PAL-003 A4 |
|----------|------------|





#### 9.1.1.3.1 Local Skin Reactions

All subjects who experience a local skin reaction during this study may be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Recommended premedications are acetaminophen and/or non-sedating antihistamine. The dosage will be standard. Because antihistamines can cause drowsiness, sedating antihistamines may be administered only if the subject is accompanied by a designated driver. Symptoms of local reactions may be treated with local application of ice and non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.2.2).

If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Sponsor's Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from study treatment.

## 9.1.1.3.2 Large Local Skin Reactions

Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be contiguous to the rAvPAL-PEG injection site, and subjects with either type of large local skin reaction may continue dosing if the skin symptoms have resolved and no other symptoms have developed. Subjects will be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses.

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

# 9.1.1.3.2.1 Large Local Skin Reactions Contiguous to Injection Site

Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may remain in the study if the skin symptoms have resolved and no other symptoms have developed. For the remainder of the study, subjects will be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable).

|----------|------------|---------|

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

#### 9.1.1.3.2.2 Large Local Skin Reactions Not Contiguous to Injection Site

Large local skin reactions that are not contiguous to the injection site may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure to rAvPAL-PEG and, therefore, will be managed as a systemic reaction (refer to Section 9.1.1.3.3). An example of a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk.

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

#### 9.1.1.3.3 Systemic Reactions

Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a definition) after administration of rAvPAL-PEG must stop further administrations of rAvPAL-PEG and must immediately return to the clinic for safety assessments. Subjects who experience generalized skin symptoms are included in this category. Immediately after the systemic reaction (within 48 hours), subjects with generalized skin symptoms must have additional assessments performed for safety (ie, Unscheduled Hypersensitivity Reaction Visit): serum antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti rAvPAL-PEG IgE, anti-rAvPAL-PEG neutralizing antibodies); serum tryptase level (it is recommended that this sample be drawn immediately after reaction); sedimentation rate; CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub>; skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction); and clinical laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1.

Following the reaction, subjects will be required to complete the assessments of the Unscheduled Hypersensitivity Reaction visit, including assessment of IgE. If a subject presents with a clinical diagnosis of anaphylaxis, further dosing will be held while laboratory evaluation of IgE, as part of the Unscheduled Systemic Reaction Visit, is performed. Subjects who do not have an IgE-mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 1 week. If laboratory data shows that the subject experienced an IgE-mediated reaction, dosing

|----------|------------|---------|

will not resume until review of the case with the Investigator, Sponsor's Medical Officer, and an allergist/immunologist.

rAvPAL-PEG administration will resume at the next lowest dose level. Restarting of rAvPAL-PEG administration following a systemic reaction must be performed in the clinic for the first week of resumed dosing. Subjects must be premedicated orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30-60 minutes following every administration of study drug. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

If blood Phe concentrations are not 60-600 µmol/L following 1 week of daily administration at the lowered dose cohort and there is no further evidence of toxicity (ie, another systemic reaction attributed to rAvPAL-PEG administration or clinically significant abnormal laboratory test results), the subject may be administered the next highest dose level in the clinic per the allowable dose increases outlined in Section 9.1.2. Subjects must be premedicated orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30-60 minutes following every study drug administration. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

#### 9.1.2 Dose Modifications

# 9.1.2.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Sponsor's Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

• The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.

|--------------------|
|--------------------|

- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg) or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject.
- The dose may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 5.0 mg/kg. Subjects who increase their dose frequency should perform the Interim Dosing Visit assessments (refer to Section 12.3.6 and Table 9.1.1).
- When a dose is increased, the subject must be observed for 30-60 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

# 9.1.2.2 Dose Decrease Methodology

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse event (any hypersensitivity reaction as defined in Section 9.1.1.2). Dose decreases may occur for safety (ie, any adverse event that may be improved with a lower, more frequent dose).

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration, dosing frequency may be reduced.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L as measured by serum Phe levels for a minimum of 1 month), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).



#### 9.1.3 Safety Assessment Criteria

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principle Investigator (PI) and the Sponsor's Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level.

# 9.1.4 Stopping Criteria

If 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate.

## 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

#### 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.

|----------|------------|---------|

- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

#### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from a previous rAvPAL-PEG study.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.



#### 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study treatment should continue to perform the study tests and evaluations until study completion. For subjects who discontinue from the study, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study treatment include, but are not limited to, the following:

- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.

If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

|-----------------------------|
|-----------------------------|

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

## 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in their previous rAvPAL-PEG study. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.

#### 9.4 Treatments

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies will be dosed with the same or higher dose that was administered upon completion of that study provided that there was no interruption in dosing. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed to by the PI and the Sponsor's Medical Officer, based upon the subject's response to doses.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects may be eligible to self administer study drug if he or she meets the following criteria:

- The subject is on a stable dosing regimen for 2 weeks (ie, the subject has demonstrated a blood Phe level within 60-600 µmol/L for a minimum of 2 consecutive weeks).
- The subject has not experienced any CTCAE Grade 3 or higher adverse event.
- The subject has not experienced any hypersensitivity reaction to rAvPAL-PEG for at least 4 weeks.
- The subject has no cognitive impairments that may increase the safety risk of self administration per the assessment of the PI.
- The subject has been approved for self administration of study drug by the Sponsor's Medical Officer.
- The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely.
- The subject has been provided with epinephrine and has been trained on when and how to administer it.

Qualified study site personnel will train each eligible subject on all procedures for self administration of study drug under the supervision of the PI. Qualified study site personnel will also be required to observe the subject prepare and perform at least 1 injection prior to allowing the subject to self administer a dose at home. The subject will see a study site nurse or home healthcare nurse in person every week or receive a telephone call from site staff to ensure that the subject continues to perform all self-administration procedures correctly, to assess adverse events, and to answer questions throughout the duration of the study. The study site nurse or home healthcare nurse will also perform the regularly scheduled assessments and procedures as outlined in Table 9.1.1 and Section 12; the subject must perform a clinic visit monthly at minimum. Training materials and other information specific to the study site personnel are provided in the Subject Self-Administration Training Materials.

Subjects who are eligible for self administration will be provided with a Subject Study Manual. Self-administration training materials will be provided in the Subject Study Manual to supplement the in-person training provided by the qualified study site personnel. The Subject Study Manual will include step-by-step instruction on the following:

- How to prepare and perform the injections of study drug safely.
- How to receive, track, store, prepare, and return both used and unused study drug.

|--------------------|
|--------------------|

- How to safely use and dispose of syringes used for injections of study drug.
- How to use a new syringe and vial every time drug is administered.
- How to care for their injection site after an injection of study drug.
- How to identify an adverse reaction and how to report this reaction to the study site.
- How and when to use epinephrine.
- Who to contact at the study site in case of an emergency.

The PI or the Sponsor's Medical Officer may request that self administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse.

Subjects who are within the target Phe range may also be permitted to convert from weight-based dosing to fixed dosing (refer to Section 9.4.4).

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site or subject with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplying the study drug to subjects who qualify for self administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites.

Information regarding supplying study drug to subjects who qualify for self administration is provided in the Subject Self-Administration Training Materials.

# 9.4.2 Identity of Investigational Product (IP)

## 9.4.2.1 Product Characteristics and Labeling

The rAvPAL-PEG drug product for SC injection is formulated and supplied as a sterile aqueous (colorless to pale yellow) solution in clear, single-use, type-1 borosilicate glass vials. Each 3 mL vial contains  $1.5 \pm 0.2$  mL to deliver either 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration) or 15 mg of rAvPAL-PEG per 1 mL (15 mg/mL protein concentration). Each vial is filled with  $1.5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Dilution instructions are provided in a separate instruction manual.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

|----------|------------|---------|

Drug product packaging will be identified with the lot number and expiration date, and will be provided in a box labeled with the study number.

## 9.4.3 Storage

IP must be stored at  $5 \pm 3^{\circ}$  C ( $41 \pm 5^{\circ}$  F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

Specific instructions for storage of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Sponsor's Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg (or 375 mg for subjects receiving a fixed dose).

For subjects receiving weight-based dosing, dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive weeks) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information presented in Table 9.4.4.1.



Table 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen

| Weight-based<br>dose (mg/kg) | Equivalent<br>fixed dose<br>(mg) | Vol for 10<br>mg/ml<br>concentration<br>(ml) | Vol for 15<br>mg/ml<br>concentration<br>(ml) |
|---|---|---|---|
| 0.03 | 2.5 | 0.25 | 0.17 |
| 0.06 | 5 | 0.5 | 0.33 |
| 0.12 | 10 | 1 | 0.67 |
| 0.25 | 20 | 2 | 1.33 |
| 0.5 | 40 | 4 | 2.67 |
| 1.0 | 75 | 7.5 | 5 |
| 2.0 | 150 | 15 | 10 |
| 3.0 | 225 | 22.5 | 15 |
| 4.0 | 300 | 30 | 20 |
| 5.0 | 375 | 37.5 | 25 |

It is preferable that the injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). The number of injections required for an individual weighing 80 kg (about 176 pounds) is provided in Table 9.4.4.2 as an example. Note this table is for example purposes only. Dosage

|----------|------------|---------|

calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff, other qualified and trained study personnel, or qualified subjects.

Information for dosing of subjects who enroll into this study after completing previous rAvPAL studies is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10.

Instructions for administration of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials.

Table 9.4.4.2: Number of Injections Required For an Individual Weighing 80 kg

| Dose Group<br>(mg/kg) | Weight<br>(kg) | Volume of Study Drug<br>(mL) <sup>a</sup> | No. of<br>Injections <sup>b</sup> |
|---|---|---|---|
| 0.001 | 80 | 0.8 | 1 |
| 0.003 | 80 | 0.6 | 1 |
| 0.01 | 80 | 0.8 | 1 |
| 0.03 | 80 | 0.2 | 1 |
| 0.06 | 80 | 0.5 | 1 |
| 0.1 | 80 | 0.8 | 1 |
| 0.3 | 80 | 2.4 | 2 |
| 0.6 | 80 | 4.8 | 2 or 3 |
| 1.0 | 80 | 8.0 | 4 |

aStudy drug is supplied at a concentration of 10 mg/mL and is then diluted by differential amounts as specified in the PAL-003 Pharmacy Manual. Volume to be injected is calculated based on a starting volume.

Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may need to be re-evaluated (refer to Section 9.4.10).

## 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

<sup>&</sup>lt;sup>b</sup>Number of injections per dose is dependent upon site policy for SC injections. The number of injections may vary at the discretion of the Investigator.



Subjects will retain the same subject number used in their previous rAvPAL-PEG study.

#### 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study.

## 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered by clinic staff or other qualified and trained study personnel.

Subjects may self administer study drug at home if approved by the Sponsor's Medical Officer and if adequate training is provided (refer to Section 9.4).

## 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the Sponsor's Medical Officer must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in a previous rAvPAL-PEG study) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior local skin reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and/or non-sedating antihistamines (refer to Section 9.1.1). If the local skin reaction worsens with a repeat 



injection (as determined by the Investigator in consultation with the Sponsor's Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior systemic reaction to rAvPAL-PEG or a PEG-containing product may participate in this study (refer to Section 9.1.1).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

## 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

#### 9.4.10 Dose Interruption and Missed Doses

Information for dosing of subjects who enroll into this study after completing previous rAvPAL\_PEG studies is provided in Section 9.1.

During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator in consultation with the Sponsor's Medical Officer. Subjects who miss more than 2 consecutive weekly doses (weekly dosing schedule) or 3 consecutive daily doses (daily dosing schedule) for whatever reason may continue participation in this study. After a dosing interruption, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects should continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 9.1.1 during any dosing interruption.

Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study treatment per discretion of the Sponsor or Investigator (refer to Section 9.3.3).

## 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific 



accounting), IP returned, and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

## 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

Subjects who qualify for self administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials).

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

#### 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer.

A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next monthly study visit. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4.

|----------|------------|---------|

#### 9.7 Efficacy and Safety Variables

#### 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

 Table 9.7.1.1: Summary of Laboratory Assessments

| | Party Responsible for | <b>Section in Protocol for</b> |
|---|---|---|
| Laboratory Assessment | <b>Performing Test</b> | Details |
| Clinical laboratory tests | Central laboratory | 9.7.6 |
| Antibody testing | BioMarin <sup>a</sup> | 9.7.5.2 |
| PK variables | BioMarin | 9.7.3 |
| Blood Phe concentrations | Central laboratory | 9.7.2.1 |
| Pregnancy test (urine) and sedimentation rate | Local laboratory | 9.7.6, 9.7.5.1 |
| Urinalysis | Central laboratory | 9.7.6 |

Phe, phenylalanine; PK, pharmacokinetic.

#### 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, including allergy history, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

#### 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



#### 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. Weight will be measured at Screening and then monthly.

## 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the Final Follow-Up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

#### **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Screening, Week 48, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

## 9.7.2 Efficacy Variable

#### 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1).

Blood Phe may be collected monthly, rather than weekly, at the discretion of the Investigator and provided that the subject meets the following criteria:

- Is receiving a stable dose of rAvPAL-PEG (defined as no dose modifications or interruptions for at least the previous 2 weeks)
- Has a stable blood Phe level (defined as Phe between 60-600 μmol/L for at least 2 consecutive weeks)

The subject may continue to have monthly, rather than weekly, blood Phe collection provided the following do not occur:

- Blood Phe measurement > 600 μmol/L
- Blood Phe measurement ≤ 30 μmol/L



If either of these conditions occurs, then that subject should return to weekly blood Phe draws until the rAvPAL-PEG dose has been adjusted and the Phe level is again within the protocol-defined target range for at least 2 weeks.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Subjects enrolled in the Substudy will have additional PK sampling performed. For subjects participating in the Substudy, PK sampling will be performed as follows:

- For subjects who are administered rAvPAL-PEG once per week, plasma PK sampling will be performed pre-dose and every 24 hours thereafter (24, 48, 72, and 96 hours if possible), and then pre-dose of the next weekly dose.
- For subjects who are administered rAvPAL-PEG two or three times per week, plasma PK sampling will be performed pre-dose and every 24 hours during the longest period between doses, when possible, and then pre-dose of the next dose.
- For subjects who are administered rAvPAL-PEG four to seven times per week, plasma PK sampling will be performed pre-dose and every 12 hours during the longest period between doses, when possible, and then pre-dose of the next dose.

See Table 9.1.2 for additional details.

BioMarin will perform the analysis.

## 9.7.4 Exploratory Efficacy Variable

Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits on a monthly basis. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each month. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator.

## 9.7.5 Safety Variables

#### 9.7.5.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 9.1.1). Female subjects with a positive serum pregnancy test at Screening do not meet eligibility criteria for enrollment.



Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

## 9.7.5.2 Antibody Testing

Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PAL IgE, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1.3.3). Immunogenicity assays will be performed at the time points indicated in the Schedule of Events (Table 9.1.1).

BioMarin will perform all anti-body testing, except for IgE antibodies, which will be assessed by a Contract Research Organization.

## 9.7.6 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All abnormal clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the abnormal result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.

Specific days for obtaining samples are provided in Table 9.1.1 and in Section 12. The scheduled clinical laboratory tests are listed in Table 9.7.6.1. A central laboratory will be used for analysis.




**Table 9.7.6.1: Clinical Laboratory Tests** 

| <b>Blood Chemistry</b> | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if |
| Alkaline | Hematocrit | Color | -applicable <sup>a</sup> |
| Phosphatase | | | |
| ALT (SGPT) | WBC count | рН | Phenylalanine |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Sedimentation rate <sup>a</sup> |
| BUN | Differential cell count | Protein | |
| Creatinine | | Glucose | |
| GGT | | Spot urine | Additional |
| | | albumin/creatinine | Unscheduled |
| | | ratio | Hypersensitivity |
| | | | Reaction Visit Tests <sup>b</sup> |
| Total protein | | Nitrite | CH50 |
| Calcium | | Urobilinogen | $C_1, C_3, C_4$ |
| Sodium | | Hemoglobin | Serum tryptase level <sup>b</sup> |
| Potassium | | Bilirubin | CRP |
| Glucose | | | |
| Uric acid | | | Complement Testing <sup>c</sup> |
| $CO_2$ | | | $C_3$ |
| Chloride | | | $C_4$ |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; C, complement; CH50, total hemolytic complement; CO2, carbon dioxide; CRP, C-reactive protein; GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.

<sup>&</sup>lt;sup>a</sup> To be performed by central laboratory. If urine pregnancy test is positive or equivocal, serum sample will be taken and assessed by a central laboratory.

|----------|------------|---------|

<sup>&</sup>lt;sup>b</sup> Perform immediately after reaction if possible.

 $<sup>^{</sup>c}$  Complement  $C_3$  and  $C_4$  to be drawn at the Screening Visit and then quarterly or as needed to resolve abnormal test results.



#### 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a subject administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment runin).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The study period during which all non-serious AEs and SAEs will be reported begins after informed consent is obtained and the first administration of study drug and continues until 4 weeks following the last administration of study drug or the last visit of the treatment period (refer to Section 12). After informed consent but prior to initiation of study treatment, only SAEs associated with any protocol-imposed interventions will be reported. The criteria for determining, and the reporting of SAEs is provided in Section 10.2.

The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or study participation is not the cause of the AE. Resolution of AEs (with dates) should be documented on the appropriate CRF page(s) and in the subject's medical record.

The Investigator responsible for the care of the subject or qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to seriousness, which is based on subject/event outcome or action criteria usually associated

|-----------------------------|
|-----------------------------|

with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the severity of each AE using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.

| Grade | Description |
|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life-<br>threatening: hospitalization or prolongation of hospitalization<br>indicated; disabling; limiting self care activities of daily<br>living (ADL) |
| 4 | Life threatening or debilitating: consequences; urgent intervention indicated <sup>b</sup> |
| 5 | Death related to AE |

Grade 4 and 5 AEs should always be reported as SAEs.

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

<sup>&</sup>lt;sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.

|----------|------------|---------|

The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably<br>Related | The administration of IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE is more likely explained by exposure to the IP than by other factors or causes. |
| | of causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).

|--------------------|
|--------------------|

#### 10.2 Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Is fatal.
- Is life threatening.
  - Note: Life-threatening refers to an event that places the subject at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires or prolongs inpatient hospitalization.
- Results in persistent or significant disability or incapacity.
- Is a congenital anomaly or birth defect in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Is an important medical event or reaction.

The reporting period for SAEs begins after informed consent is obtained, and continues until 4 weeks following the last administration of study drug or End of Treatment Visit.

All SAEs, whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form to BioMarin Pharmacovigilance (BPV). ). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the subject's medical record.

For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).



At the last scheduled visit, the Investigator should instruct each subject to report any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study treatment.

The Investigator should notify the study Sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior study treatment. The Sponsor should also be notified if the Investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that participated in this study.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

# 10.3 Pregnancy

Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up Form in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

#### **10.4** Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "...in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the


IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours.

Examples of situations that may require urgent safety measures include discovery of the following:

- Immediate need to revise the IP administration (i.e., modified dose amount or frequency not defined in protocol).
- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.

# 10.5 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the Sponsor's Medical Officer any AEs for which the issue of seriousness is unclear or questioned. Contact information for the Sponsor's Medical Officer is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone: Fax:

E-mail:

|----------|------------|---------|

## 11 APPROPRIATENESS OF MEASUREMENTS

# 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

# 11.2 Diet Diary

A 3-day diet diary will be issued to subjects for completion and will be brought to clinic on a monthly basis for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6.

|--------------------|
|--------------------|

#### 12 STUDY PROCEDURES

# 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

## 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Chest X-ray
- 12-lead ECG
- Clinical laboratory tests (including spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis)
- Complement C<sub>3</sub> and C<sub>4</sub>
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in a previous rAvPAL-PEG study, these assessments may be the same as those used for the last visit of the previous study, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week

|----------|------------|---------|

unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done daily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

## 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (postdose)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Sponsor's Medical Officer)

#### 12.3.2 Weekly Visits

Weekly visits do not require an in-clinic visit if conducted by a home healthcare professional. However, dose modifications must be performed in the clinic. Subjects must have AEs and

|--------------------|
|--------------------|

concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. For subjects on a stable dose of rAvPAL-PEG (ie, no dose change in the last 2 weeks) and have had a phenylalanine (Phe) level at or below target range (60-600 µmol/L) for 2 consecutive weeks weekly visits may be waived and replaced by a telephone call per discretion of the Investigator but monthly visits are required.

The following study activities will be performed at the weekly visits beginning with Week 2:

- Vital signs
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
  - o Blood Phe may be collected monthly, rather than weekly, if certain criteria are satisfied (refer to Section 9.7.2.1).
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Sponsor's Medical Officer)
- Weekly telephone call
  - For those subjects performing self administration and waiving (per Investigator discretion) the weekly visit (refer to Section 12.3.7).

#### 12.3.3 Substudy Visits

For subjects participating in the PK substudy, refer to Section 9.7.3 and Table 9.1.2.

#### 12.3.4 Monthly Visits (Week 4, 8, 12, etc)

Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

|--|

Beginning with Week 4, monthly visits must be performed in the clinic and consist of all weekly activities listed above in Section 12.3.2 as well as the additional study activities listed below:

- Weight
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) For safety reasons, this test must be performed prior to the chest X-ray.
- Chest x-ray (Week 48 visit only)
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.)
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Weekly telephone call
  - For those subjects performing self administration and waiving (per Investigator discretion) the weekly visit (refer to Section 12.3.7).

# 12.3.5 Quarterly Visits (Week 12, 24, 36, etc)

Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Beginning with Week 12, quarterly visits consist of all weekly (Section 12.3.2) and monthly (Section 12.3.4) activities listed above as well as the additional study activities listed below:

- Physical examination
- Complement C<sub>3</sub> and C<sub>4</sub>
- Sedimentation rate

#### **12.3.6 Interim Dosing Visit**

Subjects who increase their dose frequency during the study from 1x/week to 2x/week or daily will have additional assessments performed for 5 weeks after the subject's rAvPAL-PEG dose frequency has been increased. If the Interim Dosing Visit coincides with a weekly, monthly, or quarterly scheduled visit, the scheduled visit assessments should also be performed. The following study activities will be performed for the Interim Dosing Visit: 

| PAL-003 A4 Page 84 | BIOMARIN | PAL-003 A4 | Page 84 |
|--------------------|----------|------------|---------|
|--------------------|----------|------------|---------|

- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Administer study drug

## 12.3.7 Weekly Telephone Visit

Subjects who are administered rAvPAL-PEG at home and/or have been approved to self administered rAvPAL-PEG, should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit:

- Injection-site self inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Confirmation of drug administration

#### 12.3.8 Unscheduled Hypersensitivity Reaction Visit

Subjects who have a systemic reaction, including a generalized skin reaction, or a large local skin reaction that is not contiguous to the injection site after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 48 hours) the reaction.

- Injection-site inspection
- Clinical laboratory tests
- Sedimentation rate
- CRP, CH50, C1, C3, and C4
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies)
- Serum tryptase level
- Skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction)
- PK sample
- Assessment of AEs



#### • Concomitant medications

Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects who do not have an IgE-mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 8 weeks. If laboratory data shows that the subject experienced an IgE-mediated reaction, dosing will not resume until review of the case with the Investigator, Sponsor's Medical Officer and an allergist/immunologist (refer to Section 9.1.1.3.3).

## 12.4 Early Termination Visit

The Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug. Subjects who terminate from study treatment early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query

|--------------------|
|--------------------|

- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)

# 12.5 Final Follow-up Visit

The final follow-up (F/U) Visit will occur 1 week after the final dose of study drug.

The following study activities will be performed at the F/U Visit:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Final Follow-up Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)

|--|

## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

## 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, ECG results, and X-ray results will also be provided.

#### 14.3 Pharmacokinetic Analysis

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration  $(T_{max})$ , maximum plasma concentration  $(C_{max})$ , half life  $(t_{1/2})$ , and clearance (CL/F). Should data become available from previous rAvPAL-PEG studies that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.



## 14.3.1 Pharmacokinetic Substudy Analysis

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

# 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 60-600 µmol/L will be summarized by each scheduled time point.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis. Information regarding this exploratory analysis will be provided in the Statistical Analysis Plan.

For subjects who completed the Substudy, the effect of stopping and re-starting rAvPAL-PEG dosing on safety, blood Phe level, and immune response will be explored. Information regarding the analysis will be provided in the Statistical Analysis Plan.

# 14.5 Determination of Sample Size

Subjects who participated in previous rAvPAL-PEG studies may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

# 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.

## 14.7 Interim Analyses

Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

|--|

## 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.

|----------|------------|---------|

## 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study. Meetings of the DMC can be convened at any time at the discretion of the DMC Chair or the Sponsor's Medical Officer. The Chair will be notified by the Sponsor's Medical Officer of all SAEs and will receive summaries of other safety data as available. The DMC will review the study data as soon as it is available during the study, on a schedule defined in the DMC Charter, and offer advice on whether or not to proceed, modify or terminate study enrollment on the basis of toxicity. Details regarding the DMC membership and safety data to be reviewed by members will be provided in a charter.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.4.

|----------|------------|---------|
|----------|------------|---------|

## 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment. If the subject has followed the Investigator's instructions, BioMarin will pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures, if these costs are not covered by health insurance or another third party that usually pays these costs. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.

|--|

#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent. If an Investigator or institution refuses to allow access to subject records because of confidentiality, arrangements must be made to allow an "interview" style of data verification.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then

|-----------------------------|
|-----------------------------|

set the status of the forms, visits, and the entire casebook to locked. Upon completion of the clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.

#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.

#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (e.g., subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.

|----------|------------|---------|

## 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.

|----------|------------|---------|

#### 21 REFERENCES

Armstrong, JK, Hempel, G, Koling, S, Chan, LS et. al. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007.

Chen, AM, Scott, MD. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001.

Davis, S, Abuchowski, A, Park, YK, Davis, FF. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981.

Fisch, RO. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000.

Gamez, A, Wang, L, Sarkissian, CN, Wendt, D et. al. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007.

Ganson, NJ, Kelly, SJ, Scarlett, E, Sundy, JS et. al. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006.

Guttler, F, Azen, C, Guldberg, P, Romstad, A et. al. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003.

Harris, JM, Chess, RB. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003.

Huttenlocher, PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000.

Kaufman, S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989.

Koch, R, Hanley, W, Levy, H, Matalon, K et. al. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003.

Lapis. Long-term Correction of PKU in the Pahenu2 Mouse by Mutant and Chemically Modified Forms of Phenylalanine Ammonium Lyase. ASHG 57th Annual Meeting The American Society of Human Genetics)2007.



Lee, PJ, Lilburn, M, Baudin, J. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003.

Levy, HL. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003.

Matalon, R, Surendran, S, Matalon, KM, Tyring, S et. al. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003.

Richter, AW, Akerblom, E. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984.

Richter, AW, Akerblom, E. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983.

Rouse, B, Azen, C. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004.

Scott, MD, Murad, KL, Koumpouras, F, Talbot, M et. al. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997.

Scriver, CR, Kaufman. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-1724.

Walter, JH, White, FJ, Hall, SK, MacDonald, A et. al. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002.

Webster, R, Didier, E, Harris, P, Siegel, N et. al. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007.



#### 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.






## 24 PROTOCOL AMENDMENT TEXT REVISIONS

The following table summarizes the revisions made to the protocol and relates the changes to the appropriate rationale (see pages 2-4). Text that has been added or inserted is indicated by <u>underlined font</u>, and deleted text is indicated by <u>strikethrough font</u>.

| Section No./Title | Revision | Rationale |
|---|---|---|
| | This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205the dose finding studies (Study PAL 002 and Study PAL 004). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects. | |
| | Because rAvPAL PEG is being assessed as a long term chronic treatment for patients with PKU, there is a need to understand the effect of a temporary dosing interruption on the safety, efficacy (blood Phe), PK, and immune response. Therefore, a Substudy has been added to this study to assess the effects of stopping and re-starting rAvPAL PEG | |
| | treatment in subjects who are on a variety of rAvPAL PEG dosing regimens (dose level and frequency). Up to 10 subjects who are on a variety of dosing regimens (dose level and frequency) in this study are eligible for participation in the Substudy and will stop dosing for a period of approximately 4 weeks. During this dosing interruption, subjects will be assessed for safety, efficacy, PK, and immune response and will continue to perform the scheduled study | |
| | A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the | |
| Section 2/Synopsis, Study<br>Rationale | PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range. | 5, 6, 16 |


The exploratory objective of the study is as follows: • To assess-evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU. The Substudy objectives are as follows: To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned. • To assess the safety and tolerability of stopping and re starting rAvPAL PEG dosing in a subset of subjects with PKU. To evaluate the effect of stopping and re-starting rAvPAL PEG dosing on blood Phe concentration in a subset of subjects with PKU. • To evaluate the effect of stopping and re starting rAvPAL PEG dosing on immune response in a subset of subjects with PKU. To assess the effect of multiple doses of rAvPAL PEG on the PK profile, in particular clearance of drug, when drug is stopped in a subset of subjects with PKU who have been previously exposed to rAvPAL PEG. Section 2/Synopsis, Objectives 5, 6, 16




This is a long-term extension of <u>rAvPAL-PEG Phase 2 studies</u> the Phase 2, open label, dose finding studies, PAL 002 and PAL 004, in approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 5.0 mg/kg/week), provided no dose-limiting toxicity is observed in <u>a PAL 002 or PAL 004 previous rAvPAL-PEG study004</u>.

Only subjects who completed the protocol defined study drug regimen in PAL 002 or PAL 004a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. Subjects who enroll from PAL 002 will either continue the dose regimen that was administered upon completion of PAL 002 or start dosing at a higher dose per the dose increase instructions. Subjects who enroll from PAL 002 may start this study at a higher dose level provided there was no interruption in dosing since completion of PAL 002 and enrollment into this study. Subjects who enroll from PAL 004 will re start rAvPAL PEG dosing in this study at the same dose level and frequency as was administered upon completion of PAL 004. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration due to restarting dosing in this study. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL 002 and PAL 004 Subjects' previous subjects' rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 µmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks). Doses will be evaluated on an individual basis.

Section 2/Synopsis, Study Design and Plan

4, 6

| BION | 1AF | SIN |
|------|-----|-----|
|------|-----|-----|

| | PAL-003 Substudy | |
|---|---|---|
| | A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have | |
| | achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications | |
| | are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed. A subset of up to | |
| | 10 subjects who are already enrolled and who have consented to participate in this study will be asked to participate in a | |
| | Substudy to assess the effect that stopping and re-starting treatment with rAvPAL PEG has on safety, efficacy, PK, and | |
| | immune response. Subjects will be eligible for participation in the Substudy provided they also meet all of the PAL 003 | |
| | eligibility criteria, have been on a stable dosing regimen for approximately 4 weeks during this study, have not had any | |
| | serious adverse events reported during PAL 003, and were not enrolled in Study PAL 004. Subjects participating in the | |
| | Substudy will have rAvPAL PEG administration halted for approximately 4 weeks regardless of their dosing regimen | |
| | (dose level and frequency). rAvPAL PEG will not be administered during the dose interruption; however, subjects will | |
| | continue to perform assessments for safety, blood Phe concentration, PK, and immune response. Subjects enrolled into | |
| | the Substudy will also have additional PK sampling performed prior to the dosing interruption and during the dosing | |
| | interruption. To allow for PK sampling once dosing is stopped, subjects may be admitted to a research facility within 8 | |
| | hours of stopping dosing where they will reside for at least 24 hours. After the dosing interruption, rAvPAL PEG | |
| | administration will be re started at the same dose level and dosing frequency that was administered prior to the dosing | |
| | interruption. Upon re starting rAvPAL PEG, the first dose must be administered in the clinic and the subject must be | |
| | observed for 30 60 minutes following administration due to restarting dosing. A follow up telephone call will be made | |
| Section 2/Synopsis, Study Design | to the subject to monitor subject safety 24 hours following the return to dosing. Additional PK sampling will also be | _ |
| and Plan | performed for the first week after the dosing interruption. | 5, 6 |
| | For subjects from PAL 002 only, Aan individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For | |
| | the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile | |
| | and blood Phe concentrations. Dose increases should be performed as follows. | |
| | Only 1 dose (level or frequency) adjustment is allowed every 2 weeks. | |
| | Blood Phe levels will be measured daily for 3 days after each dose increase (fingerstick is acceptable); more | |
| Section 2/Synopsis, Dose Increase | frequent or daily blood Phe measurements may be performed. | |
| Methodology | | 2, 7 |
| | l · | 1 |

| В | 0 1111 0 | 0 | M | A | R | IN. |
|---|----------|---|---|---|---|-----|
|---|----------|---|---|---|---|-----|

| Section 2/Synopsis, Dose<br>Decrease Methodology | If the subject develops low blood Phe (as defined by a blood Phe level ≤ 30 μmol/L as measured by serum Phe levels for a minimum of 1 month), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician). | 8 |
|---|---|---|
| | Individuals eligible to participate in this study must meet all of the following criteria: 1. Must have completed participation and all protocol defined study drug in PAL 002 or PAL 004in a previous rAvPAL-PEG study. | |
| Section 2/Synopsis, Diagnosis and All Criteria for Inclusion and | <ul> <li>Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:</li> <li>4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.</li> <li>8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from PAL 002 or PAL a 004 previous rAvPAL-PEG study004.</li> </ul> | |
| Exclusion | | 11 |




rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing  $1.5 \pm 0.2$  mL to deliver <u>either 10</u> mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration) <u>or 15 mg or rAvPAL-PEG per 1 mL (15 mg/mL protein concentration)</u>. Each vial is filled with  $1.5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies PAL 002 will be dosed with the same or higher dose than the dose that was administered upon completion of that study provided that there was no interruption in dosing. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer PAL 002. Subjects enrolling from PAL 004, will be administered the same dose that was administered upon completion of PAL 004. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on onavailable information regarding a subject's blood Phe level (60-600 μmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 6120-600 μmol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the Study Sponsor's Medical Officer, based upon the subject's response to doses.

#### Fixed Dosing

Subjects who have demonstrated efficacy (ie, blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive weeks) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-daysper-week). Subjects should convert their weight-based dose using the following table:

Section 2/Synopsis, Investigational Product, Dose, Route, and Regimen

4, 16



| | | Weight-based<br>dose (mg/kg) | Equivalent<br>fixed dose (mg) | Vol for 10 mg/ml<br>concentration (ml) | Vol for 15 mg/ml<br>concentration (ml) | | |
|---|---|---|---|---|---|---|---|
| | | 0.03 | 2.5 | 0.25 | 0.17 | | |
| | | 0.06 | <u>5</u> | 0.5 | 0.33 | | |
| | | 0.12 | <u>10</u> | <u>1</u> | <u>0.67</u> | | |
| | | 0.25 | <u>20</u> | <u>2</u> | <u>1.33</u> | | |
| | | <u>0.5</u> | <u>40</u> | <u>4</u> | <u>2.67</u> | | |
| | | <u>1.0</u> | <u>75</u> | <u>7.5</u> | <u>5</u> | | |
| | | <u>2.0</u> | <u>150</u> | <u>15</u> | <u>10</u> | | |
| S 4: 2/S : - | | <u>3.0</u> | <u>225</u> | <u>22.5</u> | <u>15</u> | | |
| Section 2/Synopsis,<br>Investigational Product, Dose, | | <u>4.0</u> | <u>300</u> | <u>30</u> | <u>20</u> | | |
| Route, and Regimen | | <u>5.0</u> | <u>375</u> | <u>37.5</u> | <u>25</u> | | 4 |
| | Subjects who participated in PAL 002 or PAL 004a previous rAvPAL-PEG study may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy. | | | | | | |
| Section 2/Synopsis, Sample Size | · | | | | | 16 | |
| Section 2/Synopsis, Substudy<br>Analysis | For subjects who completed the Substudy, the effect of stopping and re starting rAvPAL PEG dosing on safety, blood Phe level, and immune responsesteady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored. | | | | 5, 6 | | |
| Section 6/Investigators and Study<br>Administrative Structure | Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), [urinalysis], and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations and urinalysis. Pharmacokinetic (PK) analysis will be performed by BioMarin. | | | | | 12 | |

| BIOMARIN | В | 0 | M | A | R | IN <sup>®</sup> |
|----------|---|---|---|---|---|-----------------|
|----------|---|---|---|---|---|-----------------|

| Section 7.2/Previous Clinical Studies | The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002, and Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience to dateas of (JAN2011) from this ongoing study and the other ongoing Phase 2 studiesy, PAL-002 and PAL-004. | 16 |
|---|---|---|
| | Currently, rAvPAL-PEG is being investigated in two three Phase 2 clinical trials (PAL-002 and PAL-004). To date (JAN2011)As of May 2012, a total of 7033 subjects have been administered rAvPAL-PEG in Study PAL 002a rAvPAL-PEG Phase 2 study and initiation and recruitment of clinical sites is underway for Study PAL 004. | |
| | Study PAL-003 (Long-Term Extension of a Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU) is an extension study of PAL-002, and PAL-004, and 165-205 (A Phase 2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate Safety, Efficacy and Tolerability of Subcutaneously Administered rAvPAL-PEG in Patients with PKU for 24 Weeks). Once subjects | |
| | have completed Study PAL 002 or PAL a p004revious rAvPAL-PEG study004, they have the option to enroll into PAL-003 and to continue to receive doses of rAvPAL-PEG for up to an additional 60 months. The protocol was amended again (28MAR2011) to increase the starting dose for Cohort 4 from 0.03 mg/kg/week to | |
| | 1.0 mg/kg/week. To date (As of JAN2011), 33 subjects have been enrolled into the study and all 10 subjects of the substudy have been dosed with 0.1 mg/kg rAvPAL-PEG. Additional information about the safety reported as of to date (JAN2011) is provided in Section 7.4.2. | |
| | Study 165-205 is a Phase 2 study using a subject-driven dose modification schema to assess safety. In addition, fixed dosing at a drug concentration of 15 mg/mL rAvPAL-PEG will be assessed. As of May 2012, enrollment of subjects is underway for this study. | |
| | In this study, subjects inwho completed a previous rAvPAL-PEG study PAL 002 and PAL 004 will continue to be administered the same rAvPAL-PEG dose that was administered in the previous studyPAL 002 or PAL 004. If the safety, PK, and blood Phe concentration results from the previous studyeither PAL 002 or PAL 004 indicate that the | |
| Section 7.2.2/Phase 2 Studies PAL-002, PAL-004, and <u>165-205</u> | appropriate level of PEGylation and dosing regimen differs from that administered in the previous studyPAL 002 or PAL 004, the PEGylation and/or dosing regimen administered in this study may change. | 15 |

| | Because rAvPAL PEG is being assessed as a long term chronic treatment for patients with PKU, there is a need to understand the effect of a temporary dosing interruption on the safety, efficacy (blood Phe), PK, and immune response. To date (JAN2011), there is limited information on the effects of a rAvPAL PEG dose interruption in subjects with PKU. Therefore, a Substudy has been added to this study to assess the effects of stopping and re starting rAvPAL PEG treatment in subjects who are on a variety of rAvPAL PEG dosing regimens (dose level and frequency). Up to 10 subjects who are on a variety of dosing regimens (dose level and frequency) in this study are eligible for participation in the Substudy and will stop dosing for a period of approximately 4 weeks. During this dosing interruption, subjects will be assessed for safety, efficacy, PK, and immune response and will continue to perform the scheduled study assessments. There is no information regarding the pharmacokinetic (PK) profile of rAvPAL PEG when blood Phe levels are at 60 600 µmol/L for subjects on a multiple dose regimen. To address this lack of information, additional PK sampling will be performed prior to the dosing interruption. Upon restarting rAvPAL PEG, PK sampling will also be performed to allow for collection of drug exposure data (area under the plasma concentration time curve [AUC] and maximum plasma concentration [C <sub>max</sub> ]), absorption rate, and clearance for subjects who have been previously exposed to rAvPAL PEG in this Substudy. This information will allow for comparisons to be performed with subjects who were naïve to previous rAvPAL PEG treatment from the Phase 1 study, PAL 001. | |
|---|---|---|
| Section 7.3/Study Rationale | have to previous 1711/12 120 deathlene from the Flase 1 study, 1712 001. | 6, 15 |
| Section 7.3/Study Rationale | A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range. This study is an extension of previous rAvPAL-PEGthethe dose finding studies(PAL 002 and PAL 004). Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects. | 5 |
| • | | 3 |
| Section 7.4/Summary of Overall Risks and Benefits | It is not expected that data from <u>previous rAvPAL-PEG studies-PAL 002 or PAL 004-will</u> change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use | 16 |

| BIOMA | ARIN |
|-------|------|
|-------|------|

| Section 7.4.2/Toxicity Due to an Immunologic Reaction | As of May 2012, a total of 70 subjects have been administered rAvPAL-PEG in the single-dose, Phase 1 study (PAL-001) and in the repeat -dosing Phase 2 studies (PAL-002, PAL-004, and PAL-003). The dose levels in the repeat-dosing studies range from 0.001 to 5.0 mg/kg/week administered in various frequencies (including 5 days a week). The most clinically significant AEs have been hypersensitivity reactions that have led to dosing interruptions and reductions. Most of the hypersensitivity reactions have been nonserious and mild-to-moderate in severity. A total of 4 SAEs have been reported in the previous rAvPAL-PEG studies. Of these 4 SAEs, 3 have been reported as related to rAvPAL-PEG. Two of the study-drug related SAEs occurred in Study PAL-001. Both of these SAEs occurred in subjects in the lower dose cohorts: an SAE of hypersensitivity reaction in a subject in the 0.001 mg/kg cohort and an SAE of anaphylactic reaction (urticaria) in a subject in the 0.01 mg/kg cohort. Neither SAE was severe or resulted in discontinuation from the study, and both of the SAEs resolved. There were no SAEs in subjects in the higher dose cohorts (0.03 mg/kg and 0.1mg/kg) in PAL-001. The third study drug-related SAE (angioedema) occurred in a subject in Study PAL-004. The fourth SAE (urticaria, dehydration) was reported as not related to study drug and occurred in a subject in Study PAL-002. There have been no reports of anaphylaxis for any subject treated with rAvPEG-PAL (as of January 2012). | 15 |
|---|---|---|
| minumorogic reaction | Subjects who have a systemic clinical reaction at any time during this study may undergo a series of assessments to | 1.0 |
| | monitor safety, including assessment of complements, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), | |
| | and IgE antibodies. Reintroduction of rAvPAL-PEG dosing after a reaction will depend on clinical assessments and | |
| | available laboratory data, such as chemistry and urine studies, to ensure that there has been no end-organ damage prior | |
| | to resuming treatment with rAvPAL-PEG. As of May 2012, antibody titers, including positive IgE titers, have not been | |
| | predictive of future clinical reactions when dosing with rAvPAL-PEG. Additionally, subjects will be premedicated to | |
| | prevent or mitigate risk of hypersensitivity reactions (refer to Section 9.1.1.3.3). | |
| | In Study PAL 001, there were 11 subjects (out of 25 subjects in the study) with skin related reactions (injection site | |
| ı | bruising, erythema, pain, rash, swelling, and urticaria) that occurred following the single administration of rAvPAL | |
| | PEG. For all of these subjects, the reactions were generalized skin reactions or injection site skin reactions that did not | |
| ı | eompromise other organs and were not life threatening. These suspected antibody mediated responses were nonserious and mild or moderate in severity. These subjects are not considered to be at significant risk for antibody mediated | |
| | reactions with injection of rAvPAL PEG during PAL 002, PAL 004, or this study; however, specific precautions for | |
| | these subjects will be taken during this study to monitor subject safety (refer to Section 9.1.1). | |
| | In Study PAL 002, 33 subjects have been dosed to date (JAN2011), including at dose levels of 2.0 mg/kg/week (or 0.4 | |
| | mg/kg/5 days a week). Most reactions reported in these subjects have been nonserious and mild or moderate in severity. | |
| | There has been 1 SAE reported to date; the event was reported as not related to treatment with study drug. There have | |
| Section 7.4.2/Toxicity Due to an | been no reports of anaphylaxis to date (JAN2011). Subjects who have a systemic reaction during this study will undergo | |
| Immunologic Reaction | a series of assessments to monitor safety, including assessment of IgE antibodies, | 1, 15 |

| <b>B</b> IOMARIN |
|------------------|
|------------------|

| Section 7.4.2/Toxicity Due to an Immunologic Reaction | , prior to determining if dosing may resume. Additionally, subjects who have systemic reactions will be premedicated and will be monitored closely for safety (refer to Section 9.1.1.3.3 for additional information regarding continued treatment of subjects with systemic reactions during the study). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.). Administration of rAvPAL-PEG may lead to anti-PEG antibody formation, and the duration of this possible effect is not known. Subjects in the Phase 2 rAvPAL-PEG studies have developed both anti-PEG IgM and anti-PEG IgG antibodies. Antibody formation This_may limit a subject's future ability to be treated with other PEG-containing (eg, Depo-Provera) or PEGylated (eg, PEG-interferon) injectable drugs. It is therefore recommended that any PEG-containing injectable drug administered to subjects after completion of this study be done under medical observation. | 15 |
|---|---|---|
| Section 7.4.2.2/Management of Allergic Reactions | In the event of an allergic reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for antibody testingimmunology studies and complement testing. This additional testing may occur up to 6 months following the final study visit. The following measures are recommended for the treatment of allergic symptoms: • Administration of oral or IV glucocorticoids • Administration of oxygen and IV fluids. • Administration of additional symptomatic treatment (eg, acetaminiophen or ibuprofen). In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. Acetaminophen or ibuprofen (5–10 mg/kg) may also be administered. An allergy and/or immunology consultation should be sought if necessary. Information regarding the management of local skin, large local skin, and systemic reactions is provided in Section 9.1.1. Detailed instructions for the management of allergic reactions are provided in the Study Reference Manual. | 1, 10, 16 |
| Section 7.4.3/Effects of Stopping and Re-Starting rAvPAL-PEG Treatment | This section has been removed. | 6 |

| BIOMARI | N |
|---------|---|
|---------|---|


The exploratory objective of the study is as follows:

• To assess-evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

- To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.
- To assess the safety and tolerability of stopping and re starting rAvPAL PEG dosing in a subset of subjects with PKU.
- To evaluate the effect of stopping and re starting rAvPAL PEG dosing on blood Phe concentration in a subset of subjects with PKU.
- To evaluate the effect of stopping and re starting rAvPAL PEG dosing on immune response in a subset of subjects with PKU.
- To assess the effect of multiple doses of rAvPAL PEG on the PK profile, in particular clearance of drug, when drug is stopped in a subset of subjects with PKU who have been previously exposed to rAvPAL PEG.

Section 8/Study Objectives

5, 6



This is a long-term extension of <u>rAvPAL-PEG Phase 2 studies</u> the Phase 2, open label, dose finding studies, <u>PAL 002</u> and <u>PAL 004</u>, in approximately 100 subjects with PKU. The doses are planned to be in the same range as those tested in PAL-002 and PAL-004 (starting at 0.001 through 5.0 mg/kg/week), provided no dose-limiting toxicity is observed in <u>a PAL 002 or PAL 004</u> previous rAvPAL-PEG study<del>004</del>.

Only subjects who completed the protocol defined study drug regimen in PAL 002 or PAL 004a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. Subjects who enroll from PAL 002 will either continue the dose regimen that was administered upon completion of PAL 002 or start dosing at a higher dose per the dose increase instructions. Subjects who enroll from PAL 002 may start this study at a higher dose level provided there was no interruption in dosing since completion of PAL 002 and enrollment into this study. Subjects who enroll from PAL 004 will re start rAvPAL PEG dosing in this study at the same dose level and frequency as was administered upon completion of PAL 004. The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administrationdue to restarting dosing in this study. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to each-clinic monthlyvisit for review with the clinical study staff.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 μmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 μmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks; refer to Section 9.4.4). Doses will be evaluated on an individual basis.

Section 9.1/Overall Study Design and Plan

6, 14, 16

| BIOMARIN | arin |
|----------|------|
|----------|------|

| | PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. PAL 002 and PAL 004 sSubjects' previous rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 µmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks; refer to Section 9.4.4). Doses will be evaluated on an individual basis. | |
|---|---|---|
| | A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed (refer to Table 9.1.2). | |
| Section 9.1/Overall Study Design and Plan | A subset of up to 10 subjects who are already enrolled and who have consented to participate in this study will be asked to participate in a Substudy to assess the effect that stopping and re starting treatment with rAvPAL PEG has on safety, efficacy, PK, and immune response. Subjects will be eligible for participation in the Substudy provided they also meet all of the PAL 003 eligibility criteria, have been on a stable dosing regimen for approximately 4 weeks during this study, have not had any serious adverse events reported during PAL 003, and were not enrolled in Study PAL 004. Subjects participating in the Substudy will have rAvPAL PEG administration halted for approximately 4 weeks regardless of their dosing regimen (dose level and frequency). rAvPAL PEG will not be administered during the dose interruption; however, subjects will continue to perform assessments for safety, blood Phe concentration, PK, and immune response. Subjects enrolled into the Substudy will also have additional PK sampling performed prior to the dosing interruption and during the dosing interruption. | 4, 5 |
| | To allow for PK sampling once dosing is stopped, subjects may be admitted to a research facility within 8 hours of stopping dosing where they will reside for at least 24 hours. After the dosing interruption, rAvPAL PEG administration will be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. Upon re-starting rAvPAL PEG, the first dose must be administered in the clinic and the subject must be observed for 30-60 minutes following administration due to restarting dosing. A follow up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Additional PK sampling will also be performed for the first week after the dosing interruption. The Schedule of Events and interim dosingPK substudy collection schedules are presented below in Table 9.1.1 and | |
| Section 9.1/Overall Study Design and Plan | <u>Table 9.1.2</u> : , Table 9.1.3 and Table 9.1.4. | 4, 5 |
| Table 9.1.1/Schedule of Events | This table has been updated to reflect changes in this amendment. | 16 |



| Table 9.1.2/PK Substudy Dosing Regimens | This table has been added for the PK Substudy. The previous Table 9.1.2 regarding interim dosing in subjects w4rho increased dose to 2x/daily has been removed. | 5, 6 |
|---|---|---|
| Table 9.1.3/Interim Dosing Visit Schedule, Subjects Whose Dose is Increased to 2x/Week | This table has been removed. | 16 |
| Section 9.1.1.1/Subjects Who<br>Have Had Previous<br>Hypersensitivity Reactions to<br>rAvPAL-PEG or a PEG-<br>containing Product | Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from a previous PAL 002 or PAL 004-rAvPAL-PEG study are excluded from participation in this study. Subjects who experienced a generalized skin rash are included in this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in PAL 002 or PAL 0a04-previous rAvPAL-PEG study are eligible to participate in this study. Subjects who have had a previous reaction and are deemed eligible for participation must be premedicated orally with acetaminophen and/or non-sedating antihistamines 1 hour 1-2 hours prior to study drug dosing for the remainder of the study. The premedication dosage will be standard | 3 |
| Section 9.1.1.3.1/Local Skin<br>Reactions | All subjects who experience a local skin reaction during this study may be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Recommended premedications are acetaminophen and/or non-sedating antihistamine. The dosage will be standard. Because antihistamines can cause drowsiness, sedating antihistamines may be administered only if the subject is accompanied by a designated driver. Subjects who have had a local skin reaction (refer to Section 9.1.1.2 for definition) after administration of rAvPAL PEG in this study may continue if the symptoms do not worsen and no other symptoms have developed but may be premedicated with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to the next dose of study drug dosing. Because antihistamines can cause drowsiness, it should be administered only if the subject is accompanied by a designated driver. | 3 |
| Section 9.1.1.3.2/Large Local<br>Skin Reactions | Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be contiguous to the rAvPAL-PEG injection site, and subjects with either type of large local skin reaction may continue dosing if the skin symptoms have resolved and no other symptoms have developed. Subjects will be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. may be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing. Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2). | 3 |

| BIOM | ARI | N. |
|------|-----|----|
|------|-----|----|

| Section 9.1.1.3.2.1/Large Local<br>Skin Reactions Contiguous to<br>Injection Site | For the remainder of the study, subjects will be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study dosesmay be premedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to the next dose of study drug. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). | 3 |
|---|---|---|
| | Following the reaction, subjects will be required to complete the assessments of the Unscheduled Hypersensitivity Reaction visit, including assessment of IgE. If a subject presents with a clinical diagnosis of anaphylaxis, further dosing will be held while laboratory evaluation of IgE, as part of the Unscheduled Systemic Reaction Visit, is performed. Subjects who do not have an IgE-mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 1 week. If laboratory data shows that the subject experienced an IgE-mediated reaction, dosing will not resume until review of the case with the Investigator, Sponsor Medical Officer, and an allergist/immunologist. | |
| Section 9.1.1.3.3/Systemic Reactions | Following completion of the Unscheduled Systemic Reaction Visit, administration of rAvPAL PEG may resume up to 1 week following the onset of the reaction if the systemic reaction is not IgE mediated and the subject's safety will not be further compromised with resumed dosing. rAvPAL-PEG administration will resume at the next lowest dose level. Restarting of rAvPAL-PEG administration following a systemic reaction must be performed in the clinic for the first week of resumed dosing. Subjects must be premedicated orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study dosespremedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing for the remainder of the study. Additionally, subjects must be closely monitored for 30-60 minutes following every administration of study drug. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable). | 3 |

| BIOM | ARIN |
|------|------|
|------|------|

| | If blood Phe concentrations are not 60-600 µmol/L following 1 week of daily administration at the lowered dose cohort and there is no further evidence of toxicity (ie, another systemic reaction attributed to rAvPAL-PEG administration or clinically significant abnormal laboratory test results), the subject may be administered the next highest dose level in the clinic per the allowable dose increases outlined in Section 9.1.2. Subjects must be premedicated orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study dosespremedicated orally with acetaminophen and/or antihistamines (standard dosage per the package insert) 1 hour prior to study drug dosing for the remainder of the study. | |
|---|---|---|
| | Additionally, subjects must be closely monitored for 30-60 minutes following every study drug administration. Because | |
| Section 9.1.1.3.3/Systemic | antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable). | |
| Reactions | | 3 |
| | For subjects from PAL 002An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows: | |
| | Only 1 dose <del>(level or frequency)</del> adjustment is allowed every 2 weeks. | |
| | Blood Phe levels will be measured daily for 3 days after each dose increase (fingerstick is acceptable); more frequent or | |
| Section 9.1.2.1/Dose Increase | daily blood Phe measurements may be performed. | |
| Methodology | | 2, 7 |
| Section 9.1.2.2/Dose Decrease | If the subject develops low blood Phe (as defined by a blood Phe level ≤ 30 µmol/L as measured by serum Phe levels for a minimum of 1 month), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician). | |
| Methodology | | 8 |
| | <ol> <li>Must have completed participation and all protocol defined study drug in PAL 002 or PAL 004in a previous<br/>rAvPAL-PEG study.</li> </ol> | |
| Section 9.3.1/Inclusion Criteria | | 11 |

| BIOMARIN | arin |
|----------|------|
|----------|------|

| | <ol> <li>A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.</li> <li>Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from a PAL 002 or PAL-previous rAvPAL-PEG study004.</li> </ol> | |
|---|---|---|
| Section 9.3.2/Exclusion Criteria | | 16 |
| Section 9.3.4/Subject<br>Identification and Replacement of<br>Subjects | Subjects will retain the same subject number assigned in <u>their previousPAL 002 or PAL rAvPAL-PEG study 004.</u> This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used. | 16 |
| | Upon enrollment into this study, subjects from <u>previous rAvPAL-PEG studies</u> <u>PAL 002</u> will be dosed with the same or higher dose that was administered upon completion of <u>PAL 002</u> that study provided that there was no interruption in <u>dosing</u> . Subjects enrolling from PAL 004, will be administered the same dose that was administered upon completion of <u>PAL 004</u> . rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects may be eligible to self administer study drug if he or she meets the following criteria: • The subject is on a stable dosing regimen for 2 weeks ( <u>ie</u> , the subject has demonstrated a blood Phe level within | |
| | 60-600 μmol/L for a minimum of 2 consecutive weeks) The patientsubject will see a study site nurse or home healthcare nurse in person every week or receive a telephone call from site staff to ensure that the subject continues to perform all self-administration procedures correctly, to assess of adverse events, and to answer questions throughout the duration of the study | |
| Section 9.4/Treatment | Subjects who are within the target Phe range may also be permitted to convert from weight-based dosing to fixed dosing (refer to Section 9.4.4). | 4, 6, 16 |

| BIOMARIN |
|----------|
|----------|

| Section 9.4.2.1/Product Characteristics and Labeling | The rAvPAL-PEG drug product for SC injection is formulated and supplied as a sterile aqueous (colorless to pale yellow) solution in clear, single-use, type-1 borosilicate glass vials. Each 3 mL vial contains $1.5 \pm 0.2$ mL to deliver either 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration) or 15 mg of rAvPAL-PEG per 1 mL (15 mg/mL protein concentration). Each vial is filled with $1.5 \pm 0.2$ mL to allow the withdrawal and delivery of up to 1 mL of the drug product. | 4 |
|---|---|---|
| | Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed by the PI and the <u>Study Sponsor's</u> Medical Officer, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg (or 375 mg for subjects receiving a fixed dose). | |
| | For subjects receiving weight-based dosing, dosage Dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage. | |
| Section 9.4.4/Directions for | Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive weeks) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information presented in Table 9.4.4.1. | |
| Administration | Table 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen | 4 |

| <b>B</b> IOMARIN | OMAR | IN |
|------------------|------|----|
|------------------|------|----|

| | | Weight-based | Equivalent | Vol for 10 mg/ml | Vol for 15 mg/ml | | |
|---|---|---|---|---|---|---|---|
| | | dose (mg/kg) | fixed dose (mg) | concentration (ml) | concentration (ml) | | |
| | | <u>0.03</u> | <u>2.5</u> | <u>0.25</u> | <u>0.17</u> | | |
| | | 0.06 | <u>5</u> | 0.5 | 0.33 | | |
| | | 0.12 | <u>10</u> | <u>1</u> | 0.67 | | |
| | | 0.25 | <u>20</u> | <u>2</u> | <u>1.33</u> | | |
| | | <u>0.5</u> | <u>40</u> | <u>4</u> | <u>2.67</u> | | |
| | | <u>1.0</u> | <u>75</u> | <u>7.5</u> | <u>5</u> | | |
| | | 2.0 | <u>150</u> | <u>15</u> | <u>10</u> | | |
| | | <u>3.0</u> | <u>225</u> | <u>22.5</u> | <u>15</u> | | |
| | | <u>4.0</u> | <u>300</u> | <u>30</u> | <u>20</u> | | |
| | | <u>5.0</u> | <u>375</u> | <u>37.5</u> | <u>25</u> | | |
| Table 9.4.4.1/ Directions for Administration | arm in Week 2, o | etc. Doses may be adn | ninistered in any of | the common SC areas ( | upper left arm in Week<br>upper arm, thigh, abdor<br>it is preferable to use b | nen). If dose | 4, 16 |
| Administration | G. 1 1 | | 1: : | 1.0.1 1 1 | . 1 | 1:0 1 1: | 4, 10 |
| Table 9.4.4.1/ Directions for Administration | Study drug will be administered by clinic staff, or other qualified and trained study personnel, or qualified subjects. Information for subjects who are participating in the Substudy and re start rAvPAL PEG dosing is provided in Section 9.1. Information for dosing of subjects who enroll into this study after completing Study PAL previous rAvPAL studies 004 is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10. | | | | 16 | | |
| | This will be an o | ppen-label study; no ra | undomization schedu | ile will be generated. | | | |
| Section 9.4.5/Method of Assigning Subjects to Treatment | | | | • | vious 04 rAvPAL-PEG | study. | |
| Groups | | | | | | | 16 |



| Section 9.4.6/Selection of Doses Used in the Study | This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study. and the ongoing study, PAL 002, to date (JAN2011). | 16 |
|---|---|---|
| | Use of any investigational product (with the exception of rAvPAL-PEG used in PAL 002 or PAL 004a previous rAvPAL-PEG study) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited. | |
| Section 9.4.8/Prior and Concomitant Medications | Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior local skin reaction to rAvPAL-PEG or a PEG-containing product will be premedicated with acetaminophen and/or non-sedating antihistamines (refer to Section 9.1.1) | 16 |
| Section 9.4.10/Dose Interruption and Missed Doses | Information for subjects who are participating in the Substudy and re start rAvPAL PEG dosing is provided in Section 9.1. Information for dosing of subjects who enroll into this study after completing Study PAL 002 or Study PAL previous rAvPAL PEG studies 004 is provided in Section 9.1. | 6, 16 |
| Section 9.6/Dietary or Other Protocol Restrictions | A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next monthly dose of study drug study visit. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4. | 14 |
| Table 9.7.1.1/Summary of Laboratory Assessments | This table has been updated to reflect changes made to this protocol amendment. | 16 |
| Section 9.7.1.3/Vital Sign<br>Measurements | Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, weight (kg), and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. Weight will be measured at Screening and then monthly. | 13 |
| Wedsdrellients | A chest X-ray will be performed at the Screening, Month 12Week 48, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health. | 13 |
| Section 9.7.1.5/Chest X-Ray | | 16 |

| BIOM | ARII | N |
|------|------|---|
|------|------|---|


Blood samples for Phe concentration measurements will be drawn at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1, Table 9.1.2: Table 9.1.3 and Table 9.1.4).

Blood Phe may be collected monthly, rather than weekly, at the discretion of the Investigator and provided that the subject meets the following criteria:

- <u>Is receiving a stable dose of rAvPAL-PEG (defined as no dose modifications or interruptions for at least the previous 2 weeks)</u>
- Has a stable blood Phe level (defined as Phe between 60-600 μmol/L for at least 2 consecutive weeks)

The subject may continue to have monthly, rather than weekly, blood Phe collection provided the following do not occur:

- Blood Phe measurement  $> 600 \mu mol/L$
- Blood Phe measurement  $\leq 30 \mu \text{mol/L}$

If either of these conditions occurs, then that subject should return to weekly blood Phe draws until the rAvPAL-PEG dose has been adjusted and the Phe level is again within the protocol-defined target range for at least 2 weeks.

In addition, after each administration of study drug, the subject will have a blood Phe measurement by fingerstick as outlined in Table 9.1.1, Table 9.1.2: , Table 9.1.3 and Table 9.1.4. This may be done by the subject at home.

Section 9.7.2.1/Blood Phenylalanine Concentrations

2, 7

| BIOM | ARII | 1 |
|------|------|---|
|------|------|---|

| | <ul> <li>Subjects enrolled in the Substudy will have additional PK sampling performed prior to the planned dosing interruption and upon re-introduction of rAvPAL PEG. For subjects participating in the Substudy, PK sampling will be performed as follows: <ul> <li>When dosing is stopped, PK sampling will be performed prior to the final dose and then postdose at 8 hours, 12 hours, 16 hours, 24 hours, 48, hours, 72 hours, 96 hours, 144 hours, 168 hours, and 216 hours.</li> </ul> </li> <li>When dosing is re-started, PK sampling will be performed predose and then postdose at 24 hours, 48 hours, 72 hours, 120 hours, and 168 hours. For subjects who are administered rAvPAL PEG once per week, plasma PK sampling will be performed pre-dose and every 24 hours thereafter (24, 48, 72, and 96 hours if possible), and then pre-dose of the next weekly dose.</li> </ul> | |
|---|---|---|
| | • For subjects who are administered rAvPAL-PEG two or three times per week, plasma PK sampling will be performed pre-dose and every 24 hours during the longest period between doses, when possible, and then pre-dose of the next dose. | |
| | <ul> <li>For subjects who are administered rAvPAL-PEG four to seven times per week, plasma PK sampling will be performed pre-dose and every 12 hours during the longest period between doses, when possible, and then pre- dose of the next dose.</li> </ul> | |
| Section 9.7.3/Pharmacokinetic Variables | See Table 9.1.2 for additional details. | 5, 6 |
| Section 9.7.4/Exploratory | Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits on a monthly basis. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each weekmonth. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator. | |
| Efficacy Variables | | 14 |

| BIOM | ARII | 1 |
|------|------|---|
|------|------|---|

| Section 12.2/Screening Visit | same as mose used for the last visit of the previous study, if they occur within 28 days from Day 1. | 1, 9, 16 |
|---|---|---|
| | For subjects who participated in PAL 002 or PAL 004, these assessments may be the same as those used for the Week 16 Visit of PAL 002 or the Week 16 visit of PAL 004a previous rAvPAL-PEG study, these assessments may be the same as those used for the last visit of the previous study, if they occur within 28 days from Day 1. | |
| | • Complement C <sub>3</sub> and C <sub>4</sub> | |
| | Clinical laboratory tests (including <u>spot urine albumin/creatinine ratio</u> , hematology, chemistry, and urinalysis) | |
| | • Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray. | |
| Section 11.2/Diet Diary | | 14 |
| | A 3-day diet diary will be issued to subjects for completion and will be brought to each-clinic on a monthly basis visit for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6. | |
| Table 9.7.6.1/Clinical Laboratory<br>Tests | This table has been updated to reflect changes in this amendment. | 16 |
| Section 9.7.6/Clinical Laboratory<br>Assessments | regarding whether or not <del>any the</del> abnormal result is clinically significant. | 16 |
| 0.0000000000000000000000000000000000000 | All <u>abnormal</u> clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment | |
| Section 9.7.5.2/Antibody Testing | BioMarin will perform theall antibody analysistesting, except for IgE antibodies, which will be assessed by a Contract Research Organization. | 16 |
| | Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG anti-PEG IgE, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1.3.3). ValidatedI-immunogenicity assays will be used perperformed at the time points indicated in the Schedule of Events (Table 9.1.1). | |

| BOMARIN |
|---------|
|---------|

| | 77. 1 1 1 1 1 1 1 1 | ı |
|---|---|---|
| | Vital signs, including weight | |
| | <ul> <li>Administer study drug (study drug may be administered on additional days during the week as determined by<br/>the Investigator, in agreement with the <u>Study Sponsor's</u> Medical Officer)</li> </ul> | |
| | <ul> <li>For subjects enrolling into this study from Study PAL 004, first dose of rAvPAL PEG must be given in the clinic setting and a telephone follow up with the subject must be performed 24 hours later to assess safety issues.</li> </ul> | |
| Section 12.3.1/Day 1 (Week 1) | | 13, 16 |
| | Weekly visits do not require an in-clinic visit if conducted by a home healthcare professional. However, dose modifications must be performed in the clinic. Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. For subjects on a stable dose of rAvPAL-PEG (ie, no dose change in the last 2 weeks) and have had a phenylalanine (Phe) level at or below target range (60-600 µmol/L) for 2 consecutive weeks weekly visits may be waived and replaced by a telephone call per discretion of the Investigator but monthly visits are required. • Vital signs, including weight • 3 day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drug.) | |
| | • For subjects participating in the Substudy, refer to Section 12.3.3. | |
| | Blood Phe and plasma tyrosine concentration | |
| | <ul> <li>Blood Phe may be collected monthly, rather than weekly, if certain criteria are satisfied (refer to<br/>Section 9.7.2.1).</li> </ul> | |
| | Weekly telephone call | |
| | <ul> <li>For those subjects performing self administration and waiving (per Investigator discretion) the<br/>weekly visit (refer to Section 12.3.7).</li> </ul> | |
| | <ul> <li>For subjects participating in the Substudy, refer to Section 12.3.3.</li> </ul> | |
| | In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by | |
| | fingerstick. This may be done by the subject at home. | 2, 6, 13, |
| Section 12.3.2/Weekly Visits | | 14 |




For subjects participating in the PK substudy, refer to Section 9.7.3 and Table 9.1.2: .on Day 1 of the Substudy (ie, final dose prior to interruption), Day 8, Day 15, Day 22, and Day 29 (ie, restart administration of study drug) for subjects participating in the Substudy:

- Physical examination
- Vital signs, including weight
- Clinical laboratory tests
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection site inspection (predose; postdose on Day 1; during weekly visit on Day 8, 15, 22; and postdose on Day 29)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3 day diet diary
- Serum anti rAvPAL PEG antibodies (anti PAL IgG, anti PAL IgM, anti PEG IgG, anti PEG IgM, and anti rAvPAL PEG neutralizing antibodies,)
- Blood Phe and plasma tyrosine concentration
  - When dosing is stopped, sampling for blood Phe assessment only will be performed prior to the final dose and then postdose at 8 hours, 12 hours, 16 hours, 24 hours, 48, hours, 72 hours, 96 hours, 144 hours, 168 hours, and 216 hours.

Section 12.3.3/Substudy Visits

5, 6

|----------|------------|----------|

| | <ul> <li>When dosing is re-started, sampling for blood Phe assessment only will be performed predose and then postdose at 24 hours, 48 hours, 72 hours, 120 hours, and 168 hours.</li> <li>For subjects participating in the Substudy, additional PK sampling will be performed upon the final dose prior to the planned dosing interruption and upon re-introduction of rAvPAL PEG. Refer to Section 9.7.3</li> </ul> | |
|---|---|---|
| | Administer study drug (Day 29 only) | |
| | For subjects participating in the Substudy, administration of rAvPAL PEG will not be performed for approximately 4 consecutive weeks regardless of their dosing regimen (dose level and frequency). After approximately 4 weeks of no dosing, rAvPAL PEG administration will be restarted at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of re administration must be given in the clinic setting, and a telephone follow up with the subject must be performed 24 hours later to assess safety issues. | |
| Section 12.3.3/Substudy Visits | | 5, 6 |

| B <sub>1</sub> OM | ARI | N |
|-------------------|-----|---|
|-------------------|-----|---|

| | Beginning with Week 4, Mmonthly visits must be performed in the clinic and consist of all weekly activities listed above in Section 12.3.2 as well as the additional and include additional activities and must be performed in the clinic. The following study activities listed below will be performed at the monthly visits beginning with Week 4: Vital signs Weight, including weight | |
|---|---|---|
| | • Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) For safety reasons, this test must be performed prior to the chest X-ray. | |
| | Chest x-ray (Month 12 Week 48 visit only) | |
| | Injection site inspection (previous and current injection site) | |
| | Assessment of AEs | |
| | Concomitant medications | |
| | Diet query | |
| | 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of study drugmonthly visit.) | |
| | • PK sample | |
| | For subjects participating in the Substudy, refer to Section 12.3.3. | |
| | Blood Phe and plasma tyrosine concentration | |
| | <ul> <li>Administer study drug (study drug may be administered on additional days during the week as determined by<br/>the Investigator, in agreement with the Study Medical Officer)</li> </ul> | |
| | Weekly telephone call | |
| Section 12.3.4/Monthly Visits (Week 4, 8, 12, etc) | <ul> <li>For those subjects performing self administration and waiving (per Investigator discretion) the<br/>weekly visit (refer to Section 12.3.7).</li> </ul> | 13, 14,<br>16 |
| (, 0, 12, 00) | → For subjects participating in the Substudy, refer to Section 12.3.3. | |
| Section 12.3.4/Monthly Visits (Week 4, 8, 12, etc) | <ul> <li>In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by<br/>fingerstick. This may be done by the subject at home.</li> </ul> | 13, 14,<br>16 |

| BIOM | IARI | N. |
|------|------|----|
|------|------|----|

| | Beginning with Week 12, Qquarterlyuarterly visits consist of all weekly(Section 12.3.2) and monthly (Section 12.3.4) activities listed above as well as the additional study activities listed below and include additional activities. The following study activities will be performed at the quarterly visits beginning with Week 12: • Vital signs, including weight • Clinical laboratory tests • Complement C <sub>3</sub> and C <sub>4</sub> • Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) | |
|---|---|---|
| | Injection site inspection (previous and current injection site) | |
| | ◆ Assessment of AEs | |
| | • Concomitant medications | |
| | Diet query | |
| | <ul> <li>3 day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next dose of<br/>study drug.)</li> </ul> | |
| | ● PK-sample | |
| | <ul> <li>For subjects participating in the Substudy, refer to Section 12.3.3.</li> </ul> | |
| | Blood Phe and plasma tyrosine concentration | |
| | <ul> <li>Serum anti-rAvPAL PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM,<br/>anti-rAvPAL PEG neutralizing antibodies)</li> </ul> | |
| | <ul> <li>Administer study drug (study drug may be administered on additional days during the week as determined by<br/>the Investigator, in agreement with the Study Medical Officer)</li> </ul> | |
| Section 12.3.5/Quarterly Visits (Week 12, 24, 35, etc) | • For subjects participating in the Substudy, refer to Section 12.3.3. | 1, 16 |
| Section 12.3.5/Quarterly Visits (Week 12, 24, 35, etc) | In addition, 3 days after each administration of study drug, the subject will have a blood Phe measurement by fingerstick. This may be done by the subject at home. | |



| | <ul> <li>Vital signs, including weight</li> </ul> | |
|---|---|---|
| | Administer study drug | |
| | Blood Phe measurement by fingerstick | |
| G .: 12.2.6/L .: D .: | This may be done by the subject at home. | |
| Section 12.3.6/Interim Dosing Visit | | 7, 16 |
| | Subjects who are administered rAvPAL-PEG at home and/or have been approved to self administered rAvPAL-PEG, should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit: | |
| | <ul> <li>Injection-site self inspection (previous and current injection site)</li> </ul> | |
| | • Assessment of AEs | |
| | Concomitant medications | |
| Section 12.3.7/Weekly Telephone | Confirmation of drug administration | |
| <u>Visit</u> | | 16 |
| Section 12.3.8/Unscheduled | <ul> <li>Perform immediately after reaction if possible.</li> </ul> | |
| Hypersensitivity Reaction Visit | | 3, 16 |
| Section 12.3.8/Unscheduled | Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects who do not have an IgE-mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 8 weeks. If laboratory data shows that the subject experienced an IgE-mediated reaction, dosing will not resume until review of the case with the Investigator, Sponsor Medical Officer and an allergist/immunologist Following completion of the Unscheduled Hypersensitivity Reaction Visit assessments, the subject may resume treatment with study drug per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. Subjects who have had an IgE mediated reaction must be discontinued from further study drug administration. Subjects who do not have an IgE mediated reaction may resume study drug administration under close monitoring; subjects must be premedicated orally with acetaminophen and/or antihistamines 1 hour prior to study drug dosing for the remainder of the study (refer to Section 9.1.1.3.3). | |
| Hypersensitivity Reaction Visit | | 3, 16 |
| ection 12.3.7/Weekly Telephone isit ection 12.3.8/Unscheduled typersensitivity Reaction Visit ection 12.3.8/Unscheduled | should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit: Injection-site self inspection (previous and current injection site) Assessment of AEs Concomitant medications Confirmation of drug administration Perform immediately after reaction if possible. Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects who do not have an IgE-mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 8 weeks. If laboratory data shows that the subject experienced an IgE-mediated reaction, dosing will not resume until review of the case with the Investigator, Sponsor Medical Officer and an allergist/immunologist Following completion of the Unscheduled Hypersensitivity Reaction Visit assessments, the subject may resume treatment with study drug per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. Subjects who have had an IgE-mediated reaction must be discontinued from further study drug administration. Subjects who do not have an IgE-mediated reaction may resume study drug administration under close monitoring; subjects must be premediated orally with acetaminophen and/or antihistamines I hour prior to study drug dosing for the remainder of the study (refer to | 16<br>3, 16 |



| Section 12.4/Early Termination | <ul> <li>Vital signs, including weight</li> <li>Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.</li> </ul> | |
|---|---|---|
| Visit | | 13, 16 |
| Section 12.5/Final Follow-up<br>Visit | Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray. | 16 |
| Section 14.3/Pharmacokinetic Analysis | Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $C_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F). Should data become available from PAL 002 or PAL 004 previous rAvPAL-PEG studies that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer. | 16 |
| Section 14.3.1/ <u>Pharmacokinetic</u><br><u>Substudy Analysis</u> | For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored. | 5 |
| Section 14.5/Determination of Sample Size | Subjects who participated in PAL 002 or PAL 004-previous rAvPAL-PEG studies may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy. | 16 |



### CLINICAL STUDY PROTOCOL

Study Title: Long-term Extension of a Phase 2, Open-Label, Dose-Finding

Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with

PKU

Protocol Number: PAL-003

Investigational Product: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis

phenylalanine ammonia lyase)

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria (PKU)

Sponsor: BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Development Phase: Phase 2

Sponsor's Responsible Medical

Officer:

, MD

, Clinical Sciences BioMarin Pharmaceutical Inc.

> 105 Digital Drive Novato, CA 94949

Duration: Up to 86 months or until study is terminated

Dose: 0.001 to a maximum weekly dose of 5.0 mg/kg or 375 mg/week

Date of Original Protocol:

October 08, 2008

Date of Amendment 1:

February 09, 2009

Date of Amendment 2:

October 30, 2009

May 04, 2011

Date of Amendment 4:

June 7, 2012

Date of Amendment 5:

February 28, 2014


May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.



### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Amendment: 5

Date: February 28, 2014

### RATIONALE AND SUMMARY OF CHANGES

The protocol for Study PAL-003 is being amended to make the following changes:

- 1. <u>Study Duration</u>: The PAL-003 study duration has been extended an additional 26 months to allow continued access to rAvPAL-PEG for subjects who do not qualify for participation in Study 165-302 and to further characterize the long-term safety and tolerability of rAvPAL-PEG in this patient population.
- 2. <u>Subject Population</u>: The study population has been revised to only include subjects who are on a stable rAvPAL-PEG dosing regimen of <70 mg/week or >350 mg/week. This study is intended to provide long-term access to rAvPAL-PEG until study termination or regulatory approval for subjects who are not eligible to transition into the pivotal, placebo-controlled, Phase 3 study, 165-302. Subjects who are on a stable rAvPAL-PEG dose regimen of ≥70 mg/week to ≤350 mg/week and do not transition to 165-302 will be withdrawn from this study.
- 3. Consultation by Sponsor's Medical Officer for Diet and Dose Modifications: Review and approval of diet and dose modifications by the sponsor's medical officer is no longer required for this study, except for dose increases > 350 mg/week. Significant modifications to dose and/or diet are not expected as subjects are generally on a stable maintenance rAvPAL-PEG dose regimen and are no longer performing dose titration.
- 4. Observation Time following Dose Increases or Dose Interruption: The observation period following an increase in rAvPAL-PEG dose or re-introduction of rAvPAL-PEG following a dose interruption has been reduced to 30 minutes as longer periods of observation is have not proven to be useful.
- 5. <u>Clinic Visits</u>: Clinic visits have been reduced from weekly to monthly because it is anticipated that rAvPAL-PEG dose adjustments will be infrequent (subjects are on a maintenance dose regimen) and to lessen patient burden. However, weekly telephone contacts will continue to be performed. Also, blood sampling for PK and immunogenicity assessments has been revised from monthly to every 12 weeks to better align with the long-term needs of this study and to lessen patient burden.

|--|

- 6. <u>Unscheduled Hypersensitivity Reaction Visit</u>: Assessments of urine/albumin creatinine ratio and urine N-methyl histamine have been added and sedimentation rate has been removed to align with the Hypersensitivity Reaction visit assessments performed in the Phase 3 studies. In addition, the window for the Hypersensitivity Reaction Visit has been changed to within 24 hours of event onset to enable timely assessment of hypersensitivity markers.
- 7. Immunogenicity Testing: Antibody testing has been clarified. Anti-PAL immunoglobulin E (IgE) testing is no longer required for this study because there has been no observed association between anti-PAL IgE and hypersensitivity reactions. Anti-PAL-PEG IgE testing will continue to be performed as part of the Hypersensitivity Reaction Visit assessments.
- 8. <u>Safety Analysis</u>: Details regarding analysis of hypersensitivity adverse events (AEs), including those that result in dose modification, have been added. Also, physical examination results and immunogenicity test results have been added to the safety analysis description.
- 9. <u>Adverse Event Reporting</u>: The pregnancy reporting period has been clarified as the time from informed consent to 4 weeks after the last dose of study drug. Also, AE reporting for events that are not resolved at the time of study completion has been revised; AE outcomes with resolution dates if applicable should be reported on the appropriate Case Report Form (CRF).
- 10. <u>Premedication</u>: Subjects who have a hypersensitivity reaction are no longer required to premedicate with acetaminophen and antihistamine for all subsequent doses of study drug. However, premedication prior to study drug administration is encouraged.
- 11. <u>Return to Dosing following Hypersensitivity Reactions</u>: Return to dosing following a hypersensitivity reaction should be based on investigator assessment in consultation with the Sponsor's Medical Officer.
- 12. <u>Pharmacokinetic Substudy</u>: The sample size for the PK Substudy has been clarified as up to 6 subjects.
- 13. <u>Investigational Product</u>: rAvPAL-PEG information has been updated to include information regarding the addition of 20-mg vials and prefilled syringes with rAvPAL-PEG.
- 14. <u>Clinical Background Information:</u> Results from the Phase 2 studies PAL-002, PAL-004, and PAL 165-205 have been updated to align with information provided in the Phase 3 studies.
- 15. <u>Schedule of Events and Study Procedures</u>: The Schedule of Events and the Study Procedures sections have been updated to reflect the changes to this amendment.
- 16. Sponsor's Medical Officer: The Medical Officer information has been updated.

|----------|------------|--------|

17. <u>Administrative Changes</u>: Additional minor changes have been made to improve clarity and consistency.

Specific revisions since the completion of the last protocol amendment (dated 07JUN2012) to the text of each section, including the Synopsis, are outlined in Section 24.

| BIOMARIN <sup>®</sup> PAL-003 A5 Page 5 |
|-----------------------------------------|
|-----------------------------------------|

### 2 SYNOPSIS

| NAME OF COMPANY BioMarin Pharmaceutical Inc. | SUMMARY TABLE Referring to Part of the | FOR NATIONAL<br>AUTHORITY USE |
|---|---|---|
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


**STUDY SITES**: Approximately 20 centers in the United States

PHASE OF DEVELOPMENT: Phase 2

### **STUDY RATIONALE:**

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-

|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

### **OBJECTIVES**:

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

### STUDY DESIGN AND PLAN:

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have


| BIOMARIN <sup>®</sup> PA | L-003 A5 Page 7 |
|--------------------------|-----------------|
|--------------------------|-----------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. | SUMMARY TABLE Referring to Part of the | FOR NATIONAL<br>AUTHORITY USE |
|---|---|---|
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. The first dose will be administered in the clinic, and the subject must be observed for 30 minutes following administration. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 μmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

A subject will continue in PAL-003 until one of the following occurs:

• The subject withdraws consent and discontinues from the study.

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- The subject is discontinued from the study at the discretion of the Investigator.
- The subject has completed the study through the Month 86 visit.
- The study is terminated.
- The study drug receives marketing authorization.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

Subjects who participate in this study will be required to transition into a Phase 3 study (165-302) if weekly doses of rAvPAL-PEG are between 70 mg/week and 350 mg/week (inclusive) provided that doses of rAvPAL-PEG have been stable (ie, no major change in dose for at least 4 weeks). Subjects who meet these criteria must be transitioned from PAL-003 to Study 165-302 provided they meet the 165-302 study eligibility criteria.

Subjects who are eligible for Study 165-302 but do not transition into 165-302 will be withdrawn from this study.

The PAL-003 study will continue until BMN-165 is approved by the Food and Drug Administration (FDA) for marketing in the United States or until the sponsor terminates further development of this drug for the treatment of PKU.

### PAL-003 Substudy

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed.

|----------------------------|
|----------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

## **Dose Modifications:**

### Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first
  modified dose administration. Subjects who increase their dose frequency do not need to be
  observed following injection of study drug if the increase in frequency does not increase the
  overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

### Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower, more

|--------------------|
|--------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

frequent dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be reduced.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

### Safety Assessment Criteria:

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Sponsor's Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level.

### **Stopping Criteria:**

If 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will be evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate.

# NUMBER OF SUBJECTS PLANNED:

Up to 100 subjects.

# DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:


|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's

|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.

- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from a previous rAvPAL-PEG study.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

# INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver 15 mg of rAvPAL-PE per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

Or

rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PE per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.



| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

| Prefilled Syringe | Volume | Concentration | Dose |
|-------------------|--------|---------------|--------|
| Sku #1 | 0.5 mL | 5 mg/mL | 2.5 mg |
| Sku #2 | 0.5 mL | 20 mg/mL | 10 mg |
| Sku #3 | 1.0 mL | 20 mg/mL | 20 mg |

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

### **Fixed Dosing**

Subjects who have demonstrated efficacy (ie, blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects should convert their weight-based dose using the following table:



NAME OF COMPANY **SUMMARY TABLE** FOR NATIONAL BioMarin Pharmaceutical Inc. Referring to Part of the **AUTHORITY USE** Dossier: 105 Digital Drive **ONLY:** Novato, CA 94949 Volume: NAME OF FINISHED PRODUCT: Page: rAvPAL-PEG (PEGylated recombinant Reference: Anabaena variabilis phenylalanine ammonia lyase) NAME OF ACTIVE INGREDIENT:

phenylalanine ammonia lyase

| Weight-based dose<br>(mg/kg) | Equivalent fixed dose (mg) | Vol for 10 mg/ml<br>concentration (ml)<br>(vial) | Vol for 15 mg/ml<br>concentration (ml)<br>(vial) <sup>a</sup> |
|---|---|---|---|
| 0.03 | 2.5 | 0.25 | 0.17 |
| 0.06 | 5 | 0.5 | 0.33 |
| 0.12 | 10 | 1 | 0.67 |
| 0.25 | 20 | 2 | 1.33 |
| 0.5 | 40 | 4 | 2.67 |
| 1.0 | 75 | 7.5 | 5 |
| 2.0 | 150 | 15 | 10 |
| 3.0 | 225 | 22.5 | 15 |
| 4.0 | 300 | 30 | 20 |
| 5.0 | 375 | 37.5 | 25 |

<sup>&</sup>lt;sup>a</sup> Applies to both 1.0 and 1.3 ml withdrawal.

# **DURATION OF TREATMENT:**

Up to 86 months.

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

# **CRITERIA FOR EVALUATION:**

# **Efficacy**:

Blood Phe concentrations will be measured.

### **Immunogenicity**:

The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG,


|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies, and anti-PEG-PAL IgE) will be assessed.

### **Safety**:

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs, ECG results, X-ray results, and laboratory test results.

### Pharmacokinetic:

Plasma concentrations of rAvPAL-PEG will be measured for subjects participating in the Substudy.

### STATISTICAL METHODS:

### Sample Size:

Subjects who participated in a previous rAvPAL-PEG study may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

### **Safety Analysis:**

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by—subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics for vital signs, physical examination results, ECG results, X-ray results, and

|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

### **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the Statistical Analysis Plan [SAP]) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

#### **Exploratory Analysis:**

Details regarding exploratory analyses will be provided in the SAP.

### **Substudy Analysis:**

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

### Pharmacokinetic Analysis:

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $t_{1/2}$ ), and clearance ( $T_{max}$ ).




# 3 TABLE OF CONTENTS

| 1 | TIT | LE PAG | ·E | 1 | | |
|---|---|---|---|---|--|--|
| 2 | SYNOPSIS | | | | | |
| 3 | TABLE OF CONTENTS | | | | | |
| 4 | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | | | | | |
| 5 | ETF | ······································ | | 25 | | |
| | 5.1 | Institut | tional Review Board or Ethics Committee | 25 | | |
| | 5.2 Ethical Conduct of Study | | | 25 | | |
| | 5.3 | Subjec | t Information and Informed Consent | 26 | | |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 27 | | |
| 7 | INTRODUCTION | | | 28 | | |
| | 7.1 Nonclinical Studies | | | 28 | | |
| | 7.2 | Previo | us Clinical Studies | 29 | | |
| | | 7.2.1 | Phase 1 Study, PAL-001 | 30 | | |
| | | 7.2.2 | Phase 2 Studies PAL-002, PAL-004, and 165-205 | 31 | | |
| | 7.3 | Study 1 | Rationale | 34 | | |
| | 7.4 Summary of Overall Risks and Benefits | | | | | |
| | | 7.4.1 | Toxicity Due to Exposure to Polyethylene Glycol (PEG) | 36 | | |
| | | 7.4.2 | Toxicity Due to an Immunologic Reaction | 36 | | |
| 8 | STUDY OBJECTIVES | | | | | |
| 9 | INV | ESTIGA | ATIONAL PLAN | 42 | | |
| | 9.1 | Overal | l Study Design and Plan | 42 | | |
| | | 9.1.1 | Management of Local and Systemic Reactions to rAvPAL-PEG | 50 | | |
| | | 9.1.2 | Dose Modifications | 55 | | |
| | | 9.1.3 | Safety Assessment Criteria. | 57 | | |
| | | 9.1.4 | Stopping Criteria | 57 | | |
| | 9.2 | Discus | sion of Study Design, Including Choice of Control Group | 57 | | |
| | 9.3 | Selecti | on of Study Population | 57 | | |
| B <sub>E</sub> O1 | MA | RI | N |
|-------------------|----|----|---|
|-------------------|----|----|---|


| | | 9.3.1 | Inclusion Criteria | 57 |
|---|---|---|---|---|
| | | 9.3.2 | Exclusion Criteria | 58 |
| | | 9.3.3 | Removal of Subjects from Treatment or Assessment | 59 |
| | | 9.3.4 | Subject Identification and Replacement of Subjects | 60 |
| | 9.4 | Treatme | ents | 60 |
| | | 9.4.1 | Treatments Administered | 62 |
| | | 9.4.2 | Identity of Investigational Product (IP) | 62 |
| | | 9.4.3 | Storage | 63 |
| | | 9.4.4 | Directions for Administration | 63 |
| | | 9.4.5 | Method of Assigning Subjects to Treatment Groups | 66 |
| | | 9.4.6 | Selection of Doses Used in the Study | 66 |
| | | 9.4.7 | Blinding | 66 |
| | | 9.4.8 | Prior and Concomitant Medications | 66 |
| | | 9.4.9 | Treatment Compliance | 67 |
| | | 9.4.10 | Dose Interruption and Missed Doses | 67 |
| | 9.5 | Investig | gational Product Accountability | 68 |
| | | 9.5.1 | Return and Disposition of Clinical Supplies | 68 |
| | 9.6 | Dietary | or Other Protocol Restrictions | 68 |
| | 9.7 | Efficacy | y and Safety Variables | 69 |
| | | 9.7.1 | Efficacy and Safety Measurements Assessed | 69 |
| | | 9.7.2 | Efficacy Variable | 70 |
| | | 9.7.3 | Pharmacokinetic Variables | 70 |
| | | 9.7.4 | Exploratory Efficacy Variable | 71 |
| | | 9.7.5 | Safety Variables | 71 |
| | | 9.7.6 | Clinical Laboratory Assessments | 72 |
| 10 | REP | ORTING | G ADVERSE EVENTS | 74 |
| | 10.1 | Adverse | e Events | 74 |
| | 10.2 | Serious | Adverse Events | 77 |
| | 10.2 | Dramar | 201/ | 75 |

| BIOM | 1AR | N |
|------|-----|---|
|------|-----|---|


| | 10.4 Urgent Safety Measures | 78 |
|----|--------------------------------------------------------------|----|
| | 10.5 BioMarin Pharmacovigilance Contact Information | 79 |
| 11 | APPROPRIATENESS OF MEASUREMENTS | 80 |
| | 11.1 Safety and Pharmacokinetics | 80 |
| | 11.2 Diet Diary | 80 |
| 12 | STUDY PROCEDURES | 81 |
| | 12.1 Prestudy | 81 |
| | 12.2 Screening Visit | 81 |
| | 12.3 Treatment Period | 81 |
| | 12.3.1 Day 1 (Week 1) | 82 |
| | 12.3.2 Weekly Telephone Visit | 83 |
| | 12.3.3 Substudy Visits | 83 |
| | 12.3.4 Monthly Visits (Week 4, 8, 12, etc) | 83 |
| | 12.3.5 Quarterly Visits (Week 12, 24, 36, etc) | 84 |
| | 12.3.6 Unscheduled Hypersensitivity Reaction Visit | 84 |
| | 12.4 Early Termination Visit | 85 |
| | 12.5 Final Follow-up Visit | 86 |
| 13 | DATA QUALITY ASSURANCE | 87 |
| 14 | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 88 |
| | 14.1 Statistical and Analytical Plans | 88 |
| | 14.2 Safety Analysis | 88 |
| | 14.3 Pharmacokinetic Analysis | 88 |
| | 14.3.1 Pharmacokinetic Substudy Analysis | 89 |
| | 14.4 Efficacy Analysis | 89 |
| | 14.5 Determination of Sample Size | 89 |
| | 14.6 Handling of Missing Data | 89 |
| | 14.7 Interim Analyses | 90 |
| | 14.8 Changes in the Conduct of the Study or Planned Analyses | 90 |
| 15 | DATA MONITORING COMMITTEE (DMC) | 01 |

|---|---|---|
| • | | |
| 16 COMPENSATION, IN | SURANCE, AND INDEMNITY | 92 |
| 17 CASE REPORT FORM | S AND SOURCE DOCUMENTS | 93 |
| 18 STUDY MONITORING | G AND AUDITING | 95 |
| 19 RETENTION OF RECO | ORDS | 96 |
| 20 USE OF INFORMATION | ON AND PUBLICATION | 97 |
| 21 REFERENCES | | 98 |
| 22 INVESTIGATOR RES | PONSIBILITIES | 100 |
| 22.1 Conduct of Study | and Protection of Human Subjects | 100 |
| 24 PROTOCOL AMENDA | MENT TEXT REVISIONS | 102 |
| LIST OF TABLES | | |
| Table 9.1.1: Schedule of E | vents | 45 |
| Table 9.1.2: PK Substudy I | Oosing Regimens | 49 |
| Table 9.4.4.1: Fixed Doses | for Subjects on Weight-Based Dose R | egimen64 |
| - | Number of Injections Required For an 80 kg | |
| Table 9.7.1.1: Summary of | Laboratory Assessments | 69 |
| Table 9.7.6.1: Clinical Lab | oratory Tests | 72 |
| LIST OF FIGURES | | |




#### 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

#### **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase

AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

 $AUC_{0-7 \text{ days}}$  area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen

°C degree Celsius

C<sub>3</sub> complement 3

C<sub>4</sub> complement 4

CBC complete blood count

CD Compact disk

CFR Code of Federal Regulations

CH50 total hemolytic complement

C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form

CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

|----------|------------|---------|

DBP diastolic blood pressure

DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up

g gram

GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure

ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IgE immunoglobulin E

IgG immunoglobulin G

IgM immunoglobulin M

IP investigational product

IRB Institutional Review Board

IV intravenous

kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

NAb neutralizing antibodies

NCI National Cancer Institute

NOAEL no observable adverse effect level

OTC over the counter

PAH phenylalanine hydroxylase

PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator

PK pharmacokinetics

PKU phenylketonuria

rAvPAL-PEG recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG

RBC red blood cell

SAE serious adverse event

SAP Statistical Analysis Plan

SBP systolic blood pressure

SC subcutaneous

SD standard deviation

SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase

SGPT serum glutamic pyruvate transaminase

US United States

WBC white blood cell

|-----------------------------|
|-----------------------------|

Definition of Terms:

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.

|----------|------------|---------|
|----------|------------|---------|

#### 5 ETHICS

#### 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

#### 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will 

|----------|------------|---------|

provide written, informed consent before any study-related tests or evaluations are performed.

#### 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR Part 50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



#### 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Pharmacovigilance Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations and urinalysis. Pharmacokinetic (PK) analysis will be performed by BioMarin.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.

|--------------------|
|--------------------|

#### 7 INTRODUCTION

A comprehensive review of PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

#### 7.1 Nonclinical Studies

The nonclinical program for rAvPAL-PEG has characterized the pharmacology, pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC route of administration. Pharmacology was assessed in the BTBR *Pah*<sup>enu2</sup> (ENU2) mouse model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to 2000 μM) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to male ENU2 mice, plasma Phe concentrations decreased from approximately 2000 μM to < 200 μM after 2 dose administrations. An attenuated reduction of blood Phe was seen between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe < 200 μM over the entire week, which continued for a total of 15 weeks.

In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a 2-4 week dose interruption and an 11-week dose interruption. Following both dose interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A similar interim attenuated response was observed with the longer dose interruption of approximately 11 weeks. In both of these assessments, no safety issues were noted upon re-starting dosing with rAvPAL-PEG (Lapis, 2007, ASHG 57th Annual Meeting).

Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No respiratory or central nervous system (CNS) effects were seen with SC administration of rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV effects of rAvPAL-PEG administered subcutaneously.

Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats and cynomolgus monkeys. The elimination half-life  $(t_{1/2})$  values of rAvPAL-PEG administered to 

| BIOMARIN <sup>®</sup> PAL-003 A5 Page 29 |
|------------------------------------------|
|------------------------------------------|

normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and 44 hours, respectively, and exhibited modest area under the plasma concentration-time curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the  $t_{1/2}$  was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum observed plasma concentration ( $C_{max}$ ), along with a long  $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) the AUC and the  $C_{max}$  are roughly linearly proportional.

Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given  $\geq 3$  mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey.

#### 7.2 Previous Clinical Studies

The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG

|----------|------------|---------|
|----------|------------|---------|

(Study PAL-002, Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience from this ongoing study and the other ongoing Phase 2 studies, PAL-002 and PAL-004.

#### 7.2.1 Phase 1 Study, PAL-001

The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations.

The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 µmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG.

Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows:

- rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg.
- For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level for these 5 subjects was 1113 μmol/L.
- Overall, no clinically significant reductions in blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, 0.01, and 0.03 mg/kg.
- For subjects who were administered rAvPAL-PEG at the 3 higher dose levels (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration levels, the calculated PK parameters were a mean  $T_{max}$  of 89-106 hours, a  $t_{1/2}$  of 46-120 hours, and an AUC<sub>0-t</sub>, and  $C_{max}$  that were proportional with dose. Drug exposure was slightly increased with increased dose.



#### 7.2.2 Phase 2 Studies PAL-002, PAL-004, and 165-205

Based on results from the Phase 1, single-dose study, the Phase 2 studies have been designed to evaluate rAvPAL-PEG at various doses and dosing regimens to safely achieve and maintain blood Phe reductions in subjects with PKU. Currently, there are three ongoing Phase 2 studies (PAL-002, PAL-004, 165-205); an overview of each study is presented in Section 7.2.2.1 (PAL-002), Section 7.2.2.2 (PAL-004), and Section 7.2.2.3 (165-205).

#### 7.2.2.1 Study PAL-002

Study PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria) was initiated in September 2009 and has completed enrollment. As of 10 September 2012, 40 subjects have been enrolled and 37 have completed the study. PAL-002 enrolled 11 previously exposed subjects from the single-dose study, PAL-001, and 29 subjects who were naïve to rAvPAL-PEG. Thirty-three of the 37 subjects who completed PAL-002 enrolled into this open-label extension study (PAL-003). Two subjects discontinued from the study due to lost to follow-up, relocation, or other reasons, and 1 subject discontinued from the study due to an AE (skin reaction).

The primary objective of this study was to evaluate the effect of multiple doses of rAvPAL-PEG (ranging from 0.001 mg/kg/week to 1.0 mg/kg/week) on blood Phe concentrations in subjects with PKU with up to 16 weeks of treatment. The secondary objectives of the study were to evaluate the safety and tolerability of SC injections of multiple doses of rAvPAL-PEG, to evaluate the immune response to rAvPAL-PEG, and to evaluate the PK profile of rAvPAL-PEG in subjects with PKU.

The PAL-002 study design consists of two parts. In Part 1, rAvPAL-PEG was administered as a once weekly fixed, low-dose induction regimen for 8 weeks. In Part 2, the rAvPAL-PEG dose was titrated upwards; subjects received adjustable dose increases for up to 8 weeks to achieve a target blood Phe concentration of 600 µmol/L. The doses and dosing schedules were revised with a series of protocol amendments to incorporate the information gained during conduct of this early, open-label, multiple-dose study.

A wide range of doses was planned for the PAL-002 study, beginning with doses as low as 0.001mg/kg/week. However, no substantial reductions in blood Phe level were observed in the majority of subjects who were administered rAvPAL-PEG in the initial four cohorts at doses of 0.001, 0.003, 0.01, and 0.03 mg/kg administered once per week. The absence of

|--------------------|
|--------------------|

appreciable Phe reduction after 16 weeks of treatment in this range of doses led to a decision to amend the study protocol to include a cohort with a higher starting dose of 0.1 mg/kg/week, which had been previously shown to decrease blood Phe levels to approximately 600 µmol/L in the single-dose, Phase 1 study (PAL-001). After the first 2 weeks of dosing at 0.1 mg/kg/week, transient Phe reduction was observed in this subset of subjects. However, this dosing regimen was accompanied by mild to moderate hypersensitivity reactions primarily after the second weekly dose, suggesting that additional exploration of dosing regimens would be required.

In summary, preliminary results from PAL-002 demonstrated that doses below 0.1 g/kg administered once per week were not effective in reducing Phe levels. While transient reduction of Phe was apparent at doses of at least 0.1 mg/kg given once per week, this dose regimen was associated with a high incidence of systemic hypersensitivity reactions, typically following the second weekly dose. Further escalation above this dose of 0.1 mg/kg/week would be required to sustain the effect on Phe levels over time. Increased doses would require spreading dose administration over several days per week, as once-weekly administration of higher doses would not be practical due to the large volume of study drug. Therefore, additional dosing regimens would need to be explored in a subsequent study (PAL-004).

Once subjects completed Study PAL-002, they were eligible to enroll into this open-label extension study, PAL-003 to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

### 7.2.2.2 Study PAL-004

PAL-004 (An Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Dose Levels of rAvPAL-PEG Administered Daily in Subjects With Phenylketonuria) was initiated in April 2011 and has completed enrollment. As of 10 September 2012, 16 subjects have been enrolled, 15 subjects have completed the study, and 15 subjects have enrolled into this study (PAL-003). One subject withdrew consent from continued participation prior to study completion. All subjects enrolled in this study were naïve to rAvPAL-PEG exposure.

The objective of this study was to determine if daily administration (defined as 5days/week) of rAvPAL-PEG at dose levels of 0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day was safe and effective in reducing and maintaining blood Phe concentrations to 600 µmol/L in subjects with PKU. The starting dose was 0.4 mg/kg, administered 5 days/week. A total of 12 subjects 

|--------------------|
|--------------------|

were added in sequence and were started on doses of 0.4, 0.2, 0.1, 0.06 mg, or 0.001/kg/day based on incoming safety data. Overall, subjects in PAL-004 who initiated treatment at higher daily doses of 0.1 to 0.4 mg/kg/day achieved immediate and substantial reduction of blood Phe levels, but dosing had to be temporarily reduced or interrupted due to the onset of systemic hypersensitivity reactions at approximately Day 10 of dosing. Phe reductions did not persist in the setting of temporary dose reduction or interruption, but Phe levels generally improved if higher dose levels were reinstated.

To prevent the onset of hypersensitivity reactions that were temporally associated with the onset of anti-drug IgM responses, an additional dosing strategy was assessed in PAL-004; 4 subjects initiated dosing at a low dose of 0.001 mg/kg/day or 0.06 mg/kg/day for 5 consecutive days and then dosing was suspended for 2 weeks. Dosing was restarted on Day 21 at the initial dose followed by dose titration to target Phe levels. Subjects administered this dosing regimen had similar efficacy, but the incidence of hypersensitivity reactions appeared to be similar to that of subjects who did not have the planned dose interruption, suggesting little advantage with this alternate induction regimen.

Experience from PAL-004 indicated that initiating daily rAvPAL-PEG dosing with relatively high daily doses was not sustainable due to the onset of hypersensitivity reactions that occurred approximately 9 to 12 days after the start of administration, nor was the alternate dosing regimen (2 week drug holiday) well tolerated or effective in Phe reduction. In addition, the daily treatment regimen did not reduce the time to achieve target blood Phe levels seen in previous studies. This study indicated that to improve tolerability, rAvPAL-PEG should be initiated with an induction period at doses substantially lower than 0.4mg/kg, followed by upward dose titration toward target Phe levels.

Once subjects completed Study PAL-004, they were eligible to enroll into this open-label extension study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

#### 7.2.2.3 Study 165-205

Study BMN 165-205 (A Phase 2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate Safety, Efficacy, and Tolerability of Subcutaneously Administered rAvPAL-PEG in Subjects With PKU for 24 Weeks) was initiated in May 2012. Data from ongoing Studies PAL-002, PAL-004, and PAL-003 suggested that a 4-week treatment course with weekly dosing at a fixed low dose (induction), followed by a weekly 2-fold, upward titration of rAvPAL-PEG to approximately 10-fold higher than the initiation dose (maximum of 375 mg/week) is 

|--------------------|
|--------------------|

effective and well tolerated. The objective of this study was to further assess this dosing regimen. Two rAvPAL-PEG dosing regimens were to be explored in this study: weekly low-dose induction (2.5 mg/week for 4 to 8 weeks), followed by a period of upward dose titration towards a target Phe level (600 µmol/L) followed by maintenance dosing at that level through the 24 week study duration (Group 1). The other dosing regimen planned for this study (Group 2) involved administration of a single bolus dose of 8 mg, followed by a treatment holiday of at least 3 weeks duration followed by resumption and escalation of study drug administration following a pattern similar to that employed in Group 1. A total of 24 subjects were enrolled into 165-205. In addition to confirming an effective, well-tolerated dose regimen, this study incorporated non-weight-based dosing, starting with dose administration once per week at a low dose (2.5mg) with gradual escalation and conversion of dose administration to 5x/week dosing for chronic maintenance therapy.

Once subjects have completed Study 165-205, they are eligible to enroll into this study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week, or into the Phase 3 study, BMN 165-302.

#### 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH. Approximately 1 in every 10,000 infants in North America is born with PKU Scriver, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan<sup>®</sup> is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation.

|----------|------------|---------|

However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. rAvPAL-PEG is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

This study is an extension of previous rAvPAL-PEG Phase 2 studies. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

#### 7.4 Summary of Overall Risks and Benefits

It is not expected that data from previous rAvPAL-PEG studies will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

#### 7.4.1 Toxicity Due to Exposure to Polyethylene Glycol (PEG)

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg rAvPAL-PEG SC. In rats, both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1).

In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

#### 7.4.2 Toxicity Due to an Immunologic Reaction

The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicit immune recognition and responses. Epitopes that play a role in the immune response may be rendered inaccessible by PEG (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylation does not eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing the immunogenicity of the molecule, it is reasonable to expect that some individuals may exhibit immune responses upon exposure to the drug. These immune responses may be clinically irrelevant, cause symptoms of various degrees, or lead to neutralization of biological activity. Subjects participating in clinical trials will be monitored closely with specific antibody titers sedimentation rates, and complete blood counts (CBCs).

As of May 2012, a total of 70 subjects have been administered rAvPAL-PEG in the single-dose, Phase 1 study (PAL-001) and in the repeat -dosing Phase 2 studies (PAL-002, PAL-004, and PAL-003). The dose levels in the repeat-dosing studies range from 0.001 to 5.0 mg/kg/week administered in various frequencies (including 5 days a week). The most clinically significant AEs have been hypersensitivity reactions that have led to dosing 

|----------|------------|---------|

interruptions and reductions. Most of the hypersensitivity reactions have been nonserious and mild-to-moderate in severity.

A total of 4 SAEs have been reported in the previous rAvPAL-PEG studies. Of these 4 SAEs, 3 have been reported as related to rAvPAL-PEG. Two of the study-drug related SAEs occurred in Study PAL-001. Both of these SAEs occurred in subjects in the lower dose cohorts: an SAE of hypersensitivity reaction in a subject in the 0.001 mg/kg cohort and an SAE of anaphylactic reaction (urticaria) in a subject in the 0.01 mg/kg cohort. Neither SAE was severe or resulted in discontinuation from the study, and both of the SAEs resolved. There were no SAEs in subjects in the higher dose cohorts (0.03 mg/kg and 0.1mg/kg) in PAL-001. The third study drug-related SAE (angioedema) occurred in a subject in Study PAL-004. The fourth SAE (urticaria, dehydration) was reported as not related to study drug and occurred in a subject in Study PAL-002. There have been no reports of anaphylaxis for any subject treated with rAvPEG-PAL (as of January 2012).

Subjects who have a systemic clinical reaction at any time during this study may undergo a series of assessments to monitor safety, including assessment of complements, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and IgE antibodies. Reintroduction of rAvPAL-PEG dosing after a reaction will depend on clinical assessments and available laboratory data, such as chemistry and urine studies, to ensure that there has been no end-organ damage prior to resuming treatment with rAvPAL-PEG. As of May 2012, antibody titers, including positive IgE titers, have not been predictive of future clinical reactions when dosing with rAvPAL-PEG. Additionally, subjects may be premedicated to prevent or mitigate risk of hypersensitivity reactions (refer to Section 9.1.1.3.3).

PEG itself is considered nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.), (Harris, 2003, Nat.Rev.Drug Discov.), however, antibodies against PEG may form when PEG is bound to compounds. (Harris, 2003, Nat.Rev.Drug Discov.), (Richter, 1983, Int.Arch.Allergy Appl.Immunol.). In some instances, development of such antibodies did not result in any significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). In some individuals, anti-PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti-PEG antibodies have been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.). Administration of rAvPAL-PEG may lead to anti-PEG antibody formation, and the duration of this possible effect is not known. Subjects in the Phase 2 rAvPAL-PEG studies have developed both anti-PEG IgM and anti-PEG IgG antibodies. Antibody formation may limit a

|----------|------------|---------|
|----------|------------|---------|

subject's future ability to be treated with other PEG-containing (eg, Depo-Provera) or PEGylated (eg, PEG-interferon) injectable drugs. It is therefore recommended that any PEG-containing injectable drug administered to subjects after completion of this study be done under medical observation.

#### 7.4.2.1 Systemic Skin Reactions

Two out of 25 subjects who were enrolled in Study PAL-001 and received the protocol-defined single dose of rAvPAL-PEG reported systemic skin reactions (generalized skin rash) that were attributed to treatment with study drug. One subject received a single dose of 0.001 mg/kg rAvPAL-PEG, and the other subject received a single dose of 0.01 mg/kg rAvPAL-PEG. One of these events was reported as serious, and the other was reported as nonserious; both events were reported following administration of Depo-Provera injections (medroxyprogesterone injection), an injectable contraception. These allergic reactions are thought to be related to the PEG molecules that are found in both the study drug, rAvPAL-PEG, and Depo-Provera. These reactions are not likely to be experienced concurrent with other birth control medications.

The 2 subjects were administered study drug during PAL-001 and then experienced an

allergic reaction following an injection of Depo-Provera. The symptoms of the reactions were hives on the arms and legs and difficulty breathing. The symptoms for both subjects resolved within 1 day following treatment with medication, including the Both subjects were examined by an allergy specialist after they completed participation in PAL-001. A skin prick test with Depo-Provera was administered as part of this examination. One subject had a mild allergic reaction to the test; however, no further reactions or complications were reported following subsequent administration of a full dose of Depo-Provera. Upon study completion, the subject continued to receive regular doses (every 3 months) of Depo-Provera, and no further reactions were reported. The second subject also had a positive reaction to Depo-Provera following administration of the skin prick test. When a subsequent full dose of Depo-Provera was administered, developed hives, itching, and chills. The subject's symptoms resolved within 1 day of taking medication prescribed by an allergist. See Section 7.2.1 for the results from Study PAL-001.

The active drug substance in rAvPAL-PEG is a bacterial protein that may elicit immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and others. The results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys indicated the formation of anti-rAvPAL antibody titers that did not correspond with observations of

the formation of anti-rAvPAL antibody titers that did not correspond with observations of injection-site reactions. Quantitation of anti-PEG titers were not assessed in the chronic repeat-dose studies in the rat and monkey. Although results from nonclincal studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys did not indicate signs of immune-mediated toxicities, it is possible that the physio-chemical properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG in humans. It is currently unknown whether administration of PEG-containing drugs, such as Depo-Provera, has a sensitizing effect to PEG in rAvPAL-PEG when administered in humans. Because the exact basis for these reported events and their duration is not known, the use of PEG-containing injectable drugs prior to, during, and after this study is prohibited as a precautionary measure (refer to Section 9.3.2 and Section 9.4.8).

#### 7.4.2.2 Management of Hypersensitivity Reactions

Hypersensitivity reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 30minutes post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of hypersensitivity reactions. Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection. Subjects who qualify for self administration of study drug will be provided with emergency resuscitation instructions (refer to Section 9.4 and the Subject Self-Administration Training Materials).

In the event of a hypersensitivity reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for immunology studies and complement testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of hypersensitivity reaction symptoms:

- Maintain the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.

|--------------------|
|--------------------|

- Administration of oral or IV glucocorticoids.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment (eg, acetaminiophen or ibuprofen).
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. An allergy and/or immunology consultation should be sought if necessary. Information regarding the management of local skin, large local skin, and systemic reactions is provided in Section 9.1.1. Detailed instructions for the management of hypersensitivity reactions are provided in the Study Reference Manual.



#### 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objective is as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

|--|

#### 9 INVESTIGATIONAL PLAN

#### 9.1 Overall Study Design and Plan

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity was observed in a previous rAvPAL-PEG studies.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the Sponsor's Medical Officer. The first dose will be administered in the clinic, and the subject must be observed for 30 minutes following administration. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to clinic monthly for review with the clinical study staff.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self administration. Additional information is provided in the Subject Self-Administration Training Materials.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003.

In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 9.1.1 and Table 9.1.2. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator.
- The subject has completed the study through the Month 86 visit.
- The study is terminated.
- The study drug receives marketing authorization.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

Subjects who participate in this study will be required to transition into a Phase 3 study (165-302) if weekly doses of rAvPAL-PEG are between 70 mg/week and 350 mg/week (inclusive) provided that doses of rAvPAL-PEG have been stable (ie, no major change in dose for at least 4 weeks). Subjects who meet these criteria must be transitioned from PAL-003 to Study 165-302 provided they meet the 165-302 study eligibility criteria.

Subjects who are eligible for Study 165-302 but do not transition into 165-302 will be withdrawn from this study.

The PAL-003 study will continue until BMN-165 is approved by the FDA for marketing in the United States or until the sponsor terminates further development of this drug for treatment of PKU.

|----------|------------|---------|

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed (refer to Table 9.1.2).

The Schedule of Events and PK substudy collection schedules are presented below in Table 9.1.1 and Table 9.1.2




### **Table 9.1.1: Schedule of Events**

| | | | Tre | atment Perio | od <sup>b,c</sup> | | | Self<br>Administration | | Unsched. |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Monthly b (eg (eg, Wk 4, Wk 12 | Quarterly<br>(eg,<br>Wk 12, 24,<br>etc.) | Visit | Final F/U<br>Visit | | Early<br>Term.<br>Visit | |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at<br>Week 2 | Every 4th week; | Every 12th<br>week.<br>Perform in<br>addition to<br>monthly<br>procedures | Up to daily | 1 week<br>after final<br>dose | | 4 weeks<br>after<br>final<br>dose | Hyper.<br>Reaction<br>Visit. <sup>d</sup><br>Perform<br>within<br>24 hours |
| Informed consent | X | | | | | | | | | |
| Medical history, including allergy history, and demographics | X | | | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | | X | | X | | X | |
| Vital signs <sup>e</sup> | X | X | | X | | X | | | X | X |
| Weight | X | | | X | | | | | | |
| 12-lead ECG | X | | | | | | X | | X | |
| Clinical laboratory tests <sup>f</sup> | X | | | X | | | X | | X | $X^g$ |
| Complements C <sub>3</sub> and C <sub>4</sub> <sup>h</sup> | X | | | | X | | | | | X |
| Sedimentation rate | | X | | | X | | X | | X | |
| Chest x-ray | X | | | X<br>(Week 48<br>visit only) | | | X | | X | |
| Urine pregnancy test <sup>i</sup> | X | X | | X | | | X | | X | |




| | | | Tre | atment Perio | od <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Monthly b (eg, Wk 4, 8, etc.) | Quarterly<br>(eg,<br>Wk 12, 24,<br>etc.) | Interim<br>Clinician<br>Visit<br>(HHRN<br>or Site) | Final F/U<br>Visit | Self<br>Administration | Early<br>Term.<br>Visit | Unsched. |
| Assessments and Events | Screeninga | D1 | Starting at<br>Week 2 | Every 4th week; | Every 12th<br>week.<br>Perform in<br>addition to<br>monthly<br>procedures | Up to<br>daily | 1 week<br>after final<br>dose | | 4 weeks<br>after<br>final<br>dose | Hyper.<br>Reaction<br>Visit. <sup>d</sup><br>Perform<br>within<br>24 hours |
| Injection-site inspectionj <sup>i j</sup> | | X<br>(postdose) | | X | | X | X | X | X | X |
| Adverse events <sup>j, k</sup> | X | X | | X | | X | X | X | X | X |
| Weekly phone call to self<br>admin participants only (to<br>assess AEs, Inj site reactions,<br>concomitant medications) | | | X | | | | | X | X | |
| Concomitant medications <sup>j</sup> | X | X | | X | | X | X | X | X | X |
| Diet query | X | X | | X | | | X | | X | |
| 3-Day diet diary <sup>1</sup> | | | | X | | | X | | X | |
| Serum antibodies <sup>m</sup> | | X | | | X | | X | | X | X |
| Plasma Phe and plasma tyrosine <sup>n</sup> | X | X | | X <sup>m</sup> | | | X | | X | |
| Urine albumin/creatinine ratio | | | | | | | | | | X |
| Urine N-methyl histamine | | | | | | | | | | X |




| | | | Tre | atment Perio | od <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Monthly b (eg, Wk 4, 8, etc.) | Quarterly<br>(eg,<br>Wk 12, 24,<br>etc.) | Interim<br>Clinician<br>Visit<br>(HHRN<br>or Site) | Final F/U<br>Visit | Self<br>Administration | Early<br>Term.<br>Visit | Unsched. |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at<br>Week 2 | Every 4th week; | Every 12th<br>week.<br>Perform in<br>addition to<br>monthly<br>procedures | Up to<br>daily | 1 week<br>after final<br>dose | | 4 weeks<br>after<br>final<br>dose | Hyper. Reaction Visit. <sup>d</sup> Perform within 24 hours |
| Plasma PK sample <sup>m</sup> | | X | | | X | | X | | X | |
| Administer study drug <sup>o</sup> | | X | | X | | X | | X | | |
| Skin biopsy (optional; affected and not affected area) | | | | | | | | | | X |
| Serum tryptase level <sup>p</sup> | | | | | | | | | | X |

AE, adverse event; C<sub>3</sub>, complement 3; C<sub>4</sub>, complement 4; CH50, total hemolytic complement; CRP, C-reactive protein; D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> A separate Screening visit for this study is required only if the time between completion of the previous rAvPAL-PEG study and enrollment into PAL-003 is greater than 28 days.

<sup>&</sup>lt;sup>b</sup> Monthly visits must be performed in the clinic.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Refer to Section 9.1.1.3.3 and Section 12.3.6.

<sup>&</sup>lt;sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.




- <sup>f</sup> Clinical laboratory tests to include spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis. Urine microscopy will be performed if any urinalysis results are positive for hematuria. Refer to Table 9.7.6.1.
- <sup>g</sup> Subjects who have a systemic reaction or a large local reaction not contiguous with the injection site should be assessed for CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub> within 24 hours of the reaction.
- <sup>h</sup>Complement C<sub>3</sub> and C<sub>4</sub> will be collected at the Screening Visit and quarterly. Additional complement testing will be performed and as needed to resolve previous abnormal test results.
- <sup>i</sup> If positive or equivocal, perform serum pregnancy test.
- <sup>j</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm).
- <sup>j</sup> Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.
- <sup>k</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug to the final study visit.
- <sup>1</sup> It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.
- <sup>m</sup> Sampling should be performed predose.
- <sup>n</sup> Samples should be drawn at least 2.5 hours after a meal. At the Investigator's discretion, blood Phe may be collected more often should more frequent monitoring of blood Phe levels be clinically warranted
- <sup>o</sup> Dosing is up to 5.0 mg/kg/week or 375 mg/week, including subjects who receive more than 1 dose/week. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may be re-evaluated.
- <sup>p</sup> Mandatory for subjects who have a systemic reaction. Take sample immediately after reaction if possible.




**Table 9.1.2: PK Substudy Dosing Regimens** 

| <b>Treatment Frequency</b> | Plasma PK Sampling | Example |
|---|---|---|
| Subjects who are administered study drug once per week | Pre-dose and every 24 hours<br>thereafter (24, 48, 72, and 96<br>hours when possible), and pre-<br>dose of the next weekly dose | If dosed on Monday: Obtain PK sample pre-dose when possible – pre-dose Monday, Tuesday, Wednesday, Thursday, Friday, and pre-dose the following Monday. No further PK substudy draws. |
| Subjects who are<br>administered study drug<br>two or three times per<br>week | Pre-dose and every 24 hours during the longest period between doses, when possible, and pre-dose of the next dose. | If dosed on Monday, Thursday, and Friday: Obtain PK sample every 24 hours during the longest period between doses: Predose Monday, Tuesday, Wednesday, and pre-dose Thursday. No further PK substudy draws. |
| Subjects who are administered study drug four to seven times per week. | Pre-dose and every 12 hours during the longest period between doses, when possible, then pre-dose of the next dose. | If dosed Monday through Friday: Obtain PK sample every 12 hours during the longest period between doses (Friday to Monday): pre-dose Friday, 12 hours post-dose Friday, Saturday (24 and 36 hours post dose), Sunday (48 and 60 hours post-dose), and pre-dose the following Monday. No further PK substudy draws. |



#### 9.1.1 Management of Local and Systemic Reactions to rAvPAL-PEG

Subjects who qualify for self administration of study drug will be provided with information and instruction with regard to management of local and systemic reactions (refer to the Subject Self-Administration Training Materials).

# 9.1.1.1 Subjects Who Have Had Previous Hypersensitivity Reactions to rAvPAL-PEG or a PEG-containing Product

Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from a previous rAvPAL-PEG study are excluded from participation in this study. Subjects who have had a previous local skin reaction to rAvPAL-PEG in a previous rAvPAL-PEG study are eligible to participate in this study. Subjects who have had a previous reaction and are deemed eligible for participation must be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing for the remainder of the study. The premedication dosage will be standard. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). Subjects may develop systemic, large local skin, or local skin reactions after enrollment in PAL-003. Refer to Section 9.1.1.2 for definitions of systemic and local skin reactions. For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.

# 9.1.1.2 Definition of Reaction and Hypersensitivity Reactions to rAvPAL-PEG Administered Subcutaneously

During Study PAL-003, subjects may experience hypersensitivity reactions to rAvPAL-PEG. The hypersensitivity reactions are defined as follows:

#### Local skin reaction:

• Skin signs or symptoms in 1 affected primary location, ie, hives, wheals, or swelling or an area of erythema, redness, induration, pain, or itching at or near the site of injection.

|----------|------------|---------|

Large local skin reaction:

• Skin signs or symptoms, ie, hives, wheals, or swelling or an area of erythema, redness, or induration with pain or itching that extends beyond the site of injection by approximately 6 inches (15 cm) and/or signs or symptoms that are not contiguous to the injection site. These may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure and, therefore, will be managed as a systemic reaction when not contiguous to the injection site.

Systemic reaction (including generalized skin symptoms):

• Skin and non-skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological; and/or a fever attributed to treatment with rAvPAL-PEG ( ≥ 100.4°F or ≥ 38°C).

For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.



PAL-003 A5



#### 9.1.1.3.1 Local Skin Reactions

All subjects who experience a local skin reaction during this study may be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Recommended premedications are acetaminophen and/or non-sedating antihistamine. The dosage will be standard. Subjects must be accompanied by a designated driver (if applicable) because antihistamines can cause drowsiness. Symptoms of local reactions may be treated with local application of ice and non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.2.2).

If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Sponsor's Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from study treatment.

#### 9.1.1.3.2 Large Local Skin Reactions

Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be contiguous to the rAvPAL-PEG injection site, and subjects with either type of large local skin reaction may continue dosing if the skin symptoms have resolved and no other symptoms have developed. Subjects will be encouraged to premedicate orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses.

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

#### 9.1.1.3.2.1 Large Local Skin Reactions Contiguous to Injection Site

Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may remain in the study if the skin symptoms have resolved and no other symptoms have developed. For the remainder of the study, subjects will be encouraged to premedicate orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable).
|----------|------------|---------|

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

### 9.1.1.3.2.2 Large Local Skin Reactions Not Contiguous to Injection Site

Large local skin reactions that are not contiguous to the injection site may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure to rAvPAL-PEG and, therefore, will be managed as a systemic reaction (refer to Section 9.1.1.3.3). An example of a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk.

Symptoms of large local skin reactions may be treated with local application of ice and topical, or IV antihistamines and/or steroids as needed (refer to Section 7.4.2.2).

## 9.1.1.3.3 Systemic Reactions

Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a definition) after administration of rAvPAL-PEG must stop further administrations of rAvPAL-PEG and must immediately return to the clinic for safety assessments. Subjects who experience generalized skin symptoms are included in this category. Immediately after the systemic reaction (within 24 hours), subjects with generalized skin symptoms must have additional assessments performed for safety (ie, Unscheduled Hypersensitivity Reaction Visit): serum antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti rAvPAL-PEG IgE, anti-rAvPAL-PEG neutralizing antibodies); serum tryptase level (it is recommended that this sample be drawn immediately after reaction); urine albumin/creatinine ratio; urine N-methyl histamine; CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub>; skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction); and clinical laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1.

Following the reaction, subjects will be required to complete the assessments of the Unscheduled Hypersensitivity Reaction visit, including assessment of IgE. If a subject presents with a clinical diagnosis of anaphylaxis, further dosing will be held while laboratory evaluation of IgE, as part of the Unscheduled Systemic Reaction Visit, is performed. Subjects may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 1 week.

rAvPAL-PEG administration will resume at the next lowest dose level. Restarting of rAvPAL-PEG administration following a systemic reaction must be performed in the clinic for the first week of resumed dosing. Subjects will be encouraged to premedicate orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30 minutes following every administration of study drug. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

If blood Phe concentrations are not 60-600 µmol/L following 1 week of daily administration at the lowered dose cohort and there is no further evidence of toxicity (ie, another systemic reaction attributed to rAvPAL-PEG administration or clinically significant abnormal laboratory test results), the subject may be administered the next highest dose level in the clinic per the allowable dose increases outlined in Section 9.1.2. Subjects will be encouraged to premedicate orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30 minutes following every study drug administration. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

#### 9.1.2 Dose Modifications

# 9.1.2.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

• The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.

|---------|
| 1 |

- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events for an individual subject. Dose increases >350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

# 9.1.2.2 Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse event (any hypersensitivity reaction as defined in Section 9.1.1.2). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower, more frequent dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be reduced.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L ), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).



## 9.1.3 Safety Assessment Criteria

If an individual subject exhibits toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Sponsor's Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level.

# 9.1.4 Stopping Criteria

If 2 or more subjects at a dose level exhibit toxicity of a treatment-emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate.

# 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

### 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.

|----------|------------|---------|

- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

#### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from a previous rAvPAL-PEG study.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

|----------|------------|---------|

#### 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study treatment should continue to perform the study tests and evaluations until study completion. For subjects who discontinue from the study, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study treatment include, but are not limited to, the following:

- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.

If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

# 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in their previous rAvPAL-PEG study. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.

### 9.4 Treatments

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies will be dosed with the same or higher dose that was administered upon completion of that study provided that there was no interruption in dosing. rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased per Investigator determination based on available information regarding a subject's blood Phe level (60-600 μmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600 μmol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects may be eligible to self administer study drug if he or she meets the following criteria:

- The subject is on a stable dosing regimen for 2 weeks (ie, the subject has demonstrated a blood Phe level within 60-600 µmol/L).
- The subject has not experienced any CTCAE Grade 3 or higher adverse event.

| PAL-003 A5 Page 61 | BIOMARIN | PAL-003 A5 | Page 61 |
|--------------------|----------|------------|---------|
|--------------------|----------|------------|---------|

- The subject has not experienced any hypersensitivity reaction to rAvPAL-PEG for at least 4 weeks.
- The subject has no cognitive impairments that may increase the safety risk of self administration per the assessment of the PI.
- The subject has been approved for self administration of study drug by the Sponsor's Medical Officer.
- The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely.
- The subject has been provided with epinephrine and has been trained on when and how to administer it.

Qualified study site personnel will train each eligible subject on all procedures for self administration of study drug under the supervision of the PI. Qualified study site personnel will also be required to observe the subject prepare and perform at least 1 injection prior to allowing the subject to self administer a dose at home. The subject will see a study site nurse or home healthcare nurse in person every week or receive a telephone call from site staff to ensure that the subject continues to perform all self-administration procedures correctly, to assess adverse events, and to answer questions throughout the duration of the study. The study site nurse or home healthcare nurse will also perform the regularly scheduled assessments and procedures as outlined in Table 9.1.1 and Section 12; the subject must perform a clinic visit monthly at minimum. Training materials and other information specific to the study site personnel are provided in the Subject Self-Administration Training Materials.

Subjects who are eligible for self administration will be provided with a Subject Study Manual. Self-administration training materials will be provided in the Subject Study Manual to supplement the in-person training provided by the qualified study site personnel. The Subject Study Manual will include step-by-step instruction on the following:

- How to prepare and perform the injections of study drug safely.
- How to receive, track, store, prepare, and return both used and unused study drug.
- How to safely use and dispose of syringes used for injections of study drug.
- How to use a new syringe and vial every time drug is administered.
- How to care for their injection site after an injection of study drug.



- How to identify an adverse reaction and how to report this reaction to the study site.
- How and when to use epinephrine.
- Who to contact at the study site in case of an emergency.

The PI or the Sponsor's Medical Officer may request that self administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse.

Subjects who are within the target Phe range may also be permitted to convert from weight-based dosing to fixed dosing (refer to Section 9.4.4).

### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site or subject with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplying the study drug to subjects who qualify for self administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites.

Information regarding supplying study drug to subjects who qualify for self administration is provided in the Subject Self-Administration Training Materials.

# 9.4.2 Identity of Investigational Product (IP)

# 9.4.2.1 Product Characteristics and Labeling

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5  $\pm$  0.2 mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5  $\pm$  0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

Or

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PE per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

|----------|------------|---------|

Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

| <b>Prefilled Syringe</b> | Volume | Concentration | Dose |
|--------------------------|--------|---------------|--------|
| Sku #1 | 0.5 mL | 5 mg/mL | 2.5 mg |
| Sku #2 | 0.5 mL | 20 mg/mL | 10 mg |
| Sku #3 | 1.0 mL | 20 mg/mL | 20 mg |

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

Drug product packaging will be identified with the lot number and expiration date, and will be provided in a box labeled with the study number.

# 9.4.3 Storage

IP must be stored at  $5 \pm 3^{\circ}$  C ( $41 \pm 5^{\circ}$  F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

Specific instructions for storage of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg (or 375 mg for subjects receiving a fixed dose).

For subjects receiving weight-based dosing, dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement

obtained at baseline or at a previous measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information presented in Table 9.4.4.1.

Table 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen

| Weight-based<br>dose (mg/kg) | Equivalent fixed dose (mg) | Vol for 10<br>mg/ml<br>concentration<br>(ml) (vial) | Vol for 15<br>mg/ml<br>concentration<br>(ml) (vial) <sup>a</sup> |
|---|---|---|---|
| 0.03 | 2.5 | 0.25 | 0.17 |
| 0.06 | 5 | 0.5 | 0.33 |
| 0.12 | 10 | 1 | 0.67 |
| 0.25 | 20 | 2 | 1.33 |
| 0.5 | 40 | 4 | 2.67 |
| 1.0 | 75 | 7.5 | 5 |
| 2.0 | 150 | 15 | 10 |
| 3.0 | 225 | 22.5 | 15 |
| 4.0 | 300 | 30 | 20 |
| 5.0 | 375 | 37.5 | 25 |

<sup>&</sup>lt;sup>a</sup> Applies to both 1.0 and 1.3 ml withdrawal.

It is preferable that the injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

|--------------------|
|--------------------|

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). The number of injections required for an individual weighing 80 kg (about 176 pounds) is provided in Table 9.4.4.2 as an example. Note this table is for example purposes only. Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff, other qualified and trained study personnel, or qualified subjects.

Information for dosing of subjects who enroll into this study after completing previous rAvPAL studies is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10.

Instructions for administration of study drug for subjects who qualify for self administration are provided in the Subject Self-Administration Training Materials.

Table 9.4.4.2: Example of Number of Injections Required For an Individual Weighing 80 kg

| Dose Group<br>(mg/kg) | Weight (kg) | Volume of Study Drug (mL) <sup>a</sup> | No. of<br>Injections <sup>b</sup> |
|---|---|---|---|
| 0.001 | 80 | 0.8 | 1 |
| 0.003 | 80 | 0.6 | 1 |
| 0.01 | 80 | 0.8 | 1 |
| 0.03 | 80 | 0.2 | 1 |
| 0.06 | 80 | 0.5 | 1 |
| 0.1 | 80 | 0.8 | 1 |
| 0.3 | 80 | 2.4 | 2 |
| 0.6 | 80 | 4.8 | 2 or 3 |
| 1.0 | 80 | 8.0 | 4 |

aStudy drug is supplied at a concentration of 10 mg/mL and is then diluted (where necessary for injection) by differential amounts as specified in the PAL-003 Pharmacy Manual. Volume to be injected is calculated based on a starting volume.

<sup>&</sup>lt;sup>b</sup>Number of injections per dose is dependent upon site policy for SC injections. The number of injections may vary at the discretion of the Investigator.



Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may need to be re-evaluated (refer to Section 9.4.10).

# 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in their previous rAvPAL-PEG study.

# 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study.

# 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered by clinic staff or other qualified and trained study personnel.

Subjects may self administer study drug at home if approved by the Sponsor's Medical Officer and if adequate training is provided (refer to Section 9.4).

#### 9.4.7 Blinding

This is an open-label study.

## 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the Sponsor's Medical Officer must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in a previous rAvPAL-PEG study) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

|-----------------------------|
|-----------------------------|

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior local skin reaction to rAvPAL-PEG or a PEG-containing product will be encouraged to be premedicate with acetaminophen and/or non-sedating antihistamines (refer to Section 9.1.1). If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Sponsor's Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior systemic reaction to rAvPAL-PEG or a PEG-containing product may participate in this study (refer to Section 9.1.1).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

### 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

# 9.4.10 Dose Interruption and Missed Doses

Information for dosing of subjects who enroll into this study after completing previous rAvPAL-PEG studies is provided in Section 9.1.

During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator. Subjects who miss more than 2 consecutive weekly doses (weekly dosing schedule) or 3 consecutive daily doses (daily dosing schedule) for whatever reason may continue participation in this study. After a dosing interruption, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first dose of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30 minutes following administration due to restarting dosing. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects should continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 9.1.1 during any dosing interruption.

|--------------------|
|--------------------|

Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study treatment per discretion of the Sponsor or Investigator (refer to Section 9.3.3).

# 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), IP returned, and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

# 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

Subjects who qualify for self administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials).

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

# 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator.

A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately 

|--------------------|
|--------------------|

prior to their next monthly study visit. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4.

# 9.7 Efficacy and Safety Variables

# 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

| Laboratory Assessment | Party Responsible for<br>Performing Test | Section in Protocol for Details |
|---|---|---|
| Clinical laboratory tests | Central laboratory | 9.7.6 |
| Antibody testing | BioMarin <sup>a</sup> | 9.7.5.2 |
| PK variables | BioMarin | 9.7.3 |
| Blood Phe concentrations | Central laboratory | 9.7.2.1 |
| Pregnancy test (urine) and sedimentation rate | Local laboratory | 9.7.6, 9.7.5.1 |
| Urinalysis | Central laboratory | 9.7.6 |

**Table 9.7.1.1: Summary of Laboratory Assessments** 

Phe, phenylalanine; PK, pharmacokinetic.

# 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, including allergy history, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

### 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

### 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. Weight will be measured at Screening and then monthly.

# 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the Final Follow-Up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

# **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Screening, Week 48, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

#### 9.7.2 Efficacy Variable

# 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn monthly, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1).

Blood Phe may be collected more often than monthly at the discretion of the Investigator should more frequent monitoring of blood Phe levels be clinically required.

A central laboratory will be used for blood Phe concentration analysis.

# 9.7.3 Pharmacokinetic Variables

Subjects enrolled in the Substudy will have additional PK sampling performed. For subjects participating in the Substudy, PK sampling will be performed as follows:

• For subjects who are administered rAvPAL-PEG once per week, plasma PK sampling will be performed pre-dose and every 24 hours thereafter (24, 48, 72, and 96 hours if possible), and then pre-dose of the next weekly dose.



- For subjects who are administered rAvPAL-PEG two or three times per week, plasma PK sampling will be performed pre-dose and every 24 hours during the longest period between doses, when possible, and then pre-dose of the next dose.
- For subjects who are administered rAvPAL-PEG four to seven times per week, plasma PK sampling will be performed pre-dose and every 12 hours during the longest period between doses, when possible, and then pre-dose of the next dose.

See Table 9.1.2 for additional details.

BioMarin will perform the analysis.

# 9.7.4 Exploratory Efficacy Variable

Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits on a monthly basis. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each month. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator.

# 9.7.5 Safety Variables

#### 9.7.5.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 9.1.1). Female subjects with a positive serum pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.4 for details on the reporting procedures to follow in the event of pregnancy.

# 9.7.5.2 Antibody Testing

Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to



Section 9.1.1.3.3). Immunogenicity assays will be performed at the time points indicated in the Schedule of Events (Table 9.1.1).

BioMarin will perform all anti-body testing, except for IgE antibodies, which will be assessed by a Contract Research Organization.

# 9.7.6 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All abnormal clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the abnormal result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.

**Table 9.7.6.1: Clinical Laboratory Tests** 

| <b>Blood Chemistry</b> | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if |
| Alkaline<br>Phosphatase | Hematocrit | Color | applicable <sup>a</sup> |
| ALT (SGPT) | WBC count | рН | Phenylalanine |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Sedimentation rate <sup>a</sup> |
| BUN | Differential cell count | Protein | |
| Creatinine | | Glucose | |
| GGT | | Spot urine<br>albumin/creatinine<br>ratio | Additional Unscheduled Hypersensitivity Reaction Visit Tests <sup>b</sup> |
| Total protein | | Nitrite | CH50 |
| Calcium | | Urobilinogen | $C_1, C_3, C_4$ |
| Sodium | | Hemoglobin | Serum tryptase level <sup>b</sup> |



| <b>Blood Chemistry</b> | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Potassium | | Bilirubin | CRP |
| Glucose | | | Urine N-methyl histamine |
| | | | Urine albumin/creatinine ratio |
| Uric acid | | | Complement Testing <sup>c</sup> |
| CO <sub>2</sub> | | | C <sub>3</sub> |
| Chloride | | | C <sub>4</sub> |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; C, complement; CH50, total hemolytic complement; CO2, carbon dioxide; CRP, C-reactive protein; GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.

<sup>&</sup>lt;sup>a</sup> To be performed by central laboratory. If urine pregnancy test is positive or equivocal, serum sample will be taken and assessed by a central laboratory.

<sup>&</sup>lt;sup>b</sup> Perform immediately after reaction if possible.

<sup>&</sup>lt;sup>c</sup> Complement C<sub>3</sub> and C<sub>4</sub> to be drawn at the Screening Visit and then quarterly or as needed to resolve abnormal test results.



#### 10 REPORTING ADVERSE EVENTS

#### **10.1** Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a subject administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment runin).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The study period during which all non-serious AEs and SAEs will be reported begins after informed consent is obtained and the first administration of study drug and continues until 4 weeks following the last administration of study drug or the last visit of the treatment period (refer to Section 12). After informed consent but prior to initiation of study treatment, only SAEs associated with any protocol-imposed interventions will be reported. The criteria for determining, and the reporting of SAEs is provided in Section 10.2.

The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or study participation is not the cause of the AE. Outcome of AEs (and resolution dates) should be documented on the appropriate CRF page(s) and in the subject's medical record unless the subject is lost to follow-up or it has been determined that the study treatment or study participation is not the cause of the AE.

The Investigator responsible for the care of the subject or qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to 



seriousness, which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the severity of each AE using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.

| Grade | Description |
|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life-<br>threatening: hospitalization or prolongation of hospitalization<br>indicated; disabling; limiting self care activities of daily<br>living (ADL) |
| 4 | Life threatening or debilitating: consequences; urgent intervention indicated <sup>b</sup> |
| 5 | Death related to AE |

Grade 4 and 5 AEs should always be reported as SAEs.

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

<sup>&</sup>lt;sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.

|----------|------------|---------|

The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably<br>Related | The administration of IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE is more likely explained by exposure to the IP than by other factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).

|--------------------|
|--------------------|

#### 10.2 Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Is fatal.
- Is life threatening.
  - Note: Life-threatening refers to an event that places the subject at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires or prolongs inpatient hospitalization.
- Results in persistent or significant disability or incapacity.
- Is a congenital anomaly or birth defect in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Is an important medical event or reaction.

The reporting period for SAEs begins after informed consent is obtained, and continues until 4 weeks following the last administration of study drug or End of Treatment Visit.

All SAEs, whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form to BioMarin Pharmacovigilance (BPV). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the subject's medical record.

For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).

|----------|------------|---------|
|----------|------------|---------|

At the last scheduled visit, the Investigator should instruct each subject to report any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study treatment.

The Investigator should notify the study Sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior study treatment. The Sponsor should also be notified if the Investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that participated in this study.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

# 10.3 Pregnancy

Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. The reporting period for pregnancies begins with informed consent and continues until 4 weeks following the last study drug dose. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution to BPV in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

# **10.4** Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "...in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the



competent authorities of those new events and the measures taken and shall ensure that the IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours.

Examples of situations that may require urgent safety measures include discovery of the following:

- Immediate need to revise the IP administration (i.e., modified dose amount or frequency not defined in protocol).
- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.

# 10.5 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the Sponsor's Medical Officer any AEs for which the issue of seriousness is unclear or questioned. Contact information for the Sponsor's Medical Officer is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:
Fax:
E-mail:



#### 11 APPROPRIATENESS OF MEASUREMENTS

# 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

# 11.2 Diet Diary

A 3-day diet diary will be issued to subjects for completion and will be brought to clinic on a monthly basis for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6.

|--------------------|
|--------------------|

#### 12 STUDY PROCEDURES

# 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

# 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Chest X-ray
- 12-lead ECG
- Clinical laboratory tests (including spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis)
- Complement C<sub>3</sub> and C<sub>4</sub>
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in a previous rAvPAL-PEG study, these assessments may be the same as those used for the last visit of the previous study, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week

|--|

unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done daily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

# 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Injection-site inspection (postdose)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator)

|--|

## 12.3.2 Weekly Telephone Visit

Subjects should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit:

- Injection-site self inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Confirmation of dose level, frequency, and study drug administration

### 12.3.3 Substudy Visits

For subjects participating in the PK substudy, refer to Section 9.7.3 and Table 9.1.2.

## 12.3.4 Monthly Visits (Week 4, 8, 12, etc)

Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Beginning with Week 4, monthly visits must be performed in the clinic. The following study activities will be performed:

- Vital signs
- Weight
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) For safety reasons, this test must be performed prior to the chest X-ray.
- Chest x-ray (Week 48 visit only)
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

|----------|------------|---------|

• 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.)

## 12.3.5 Quarterly Visits (Week 12, 24, 36, etc)

Subjects must have AEs and concomitant medications assessed and an injection-site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Beginning with Week 12, quarterly visits consist of all monthly (Section 12.3.4) activities listed above as well as the additional study activities listed below:

- Physical examination
- Complement C<sub>3</sub> and C<sub>4</sub>
- Sedimentation rate
- PK sample
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)

# 12.3.6 Unscheduled Hypersensitivity Reaction Visit

Subjects who have a systemic reaction, including a generalized skin reaction, or a large local skin reaction that is not contiguous to the injection site after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 24 hours) the reaction.

- Vital signs
- Injection-site inspection
- Clinical laboratory tests
- Urine/albumin creatinine ratio
- CRP, CH50, C1, C3, and C4
- Urine N-methyl histamine
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies)

|-----------------------------|
|-----------------------------|

- Serum tryptase level
- Skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction)
- Assessment of AEs
- Concomitant medications

Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 8 weeks.

#### 12.4 Early Termination Visit

The Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug. Subjects who terminate from study treatment early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications

|--------------------|
|--------------------|

- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)

# 12.5 Final Follow-up Visit

The final follow-up (F/U) Visit will occur 1 week after the final dose of study drug.

The following study activities will be performed at the F/U Visit:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Injection-site inspection (previous injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Final Follow-up Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)

|--|

## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

# 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

# 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF).

The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics of vital signs, physical examination results, ECG results, and X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

### 14.3 Pharmacokinetic Analysis

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration 

|--|

 $(T_{max})$ , maximum plasma concentration  $(C_{max})$ , half life  $(t_{1/2})$ , and clearance (CL/F). Should data become available from previous rAvPAL-PEG studies that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the Sponsor's Medical Officer.

# 14.3.1 Pharmacokinetic Substudy Analysis

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

# 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the SAP) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis.

Details regarding exploratory analyses will be provided in the Statistical Analysis Plan.

# **14.5** Determination of Sample Size

Subjects who participated in previous rAvPAL-PEG studies may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

# 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.


## 14.7 Interim Analyses

Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

## 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.

|----------|------------|---------|

## 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Assess the effect and relevance of new external evidence.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.4.
- Make recommendations to the BioMarin concerning continuation or termination of the study or other study modifications based on observations.

|----------|------------|---------|

## 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment, unless the executed Clinical Trial Agreement between BioMarin and the institution of the investigator specifies otherwise. If the subject has followed the Investigator's instructions, BioMarin may pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.

|----------|------------|---------|

#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the

|--------------------|
|--------------------|

clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.

|--|

#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.

|--|

#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (e.g., subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.

|----------|------------|---------|
|----------|------------|---------|

## 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.

|--------------------|
|--------------------|

#### 21 REFERENCES

Armstrong, JK, Hempel, G, Koling, S, Chan, LS et. al. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007.

Chen, AM, Scott, MD. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001.

Davis, S, Abuchowski, A, Park, YK, Davis, FF. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981.

Fisch, RO. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000.

Gamez, A, Wang, L, Sarkissian, CN, Wendt, D et. al. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007.

Ganson, NJ, Kelly, SJ, Scarlett, E, Sundy, JS et. al. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006.

Guttler, F, Azen, C, Guldberg, P, Romstad, A et. al. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003.

Harris, JM, Chess, RB. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003.

Huttenlocher, PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000.

Kaufman, S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989.

Koch, R, Hanley, W, Levy, H, Matalon, K et. al. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003.

Lapis. Long-term Correction of PKU in the Pahenu2 Mouse by Mutant and Chemically Modified Forms of Phenylalanine Ammonium Lyase. ASHG 57th Annual Meeting The American Society of Human Genetics)2007.




Lee, PJ, Lilburn, M, Baudin, J. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003.

Levy, HL. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003.

Matalon, R, Surendran, S, Matalon, KM, Tyring, S et. al. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003.

Richter, AW, Akerblom, E. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983.

Richter, AW, Akerblom, E. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984.

Rouse, B, Azen, C. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004.

Scott, MD, Murad, KL, Koumpouras, F, Talbot, M et. al. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997.

Scriver, CR, Kaufman. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-1724.

Walter, JH, White, FJ, Hall, SK, MacDonald, A et. al. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002.

Webster, R, Didier, E, Harris, P, Siegel, N et. al. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007.



#### 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.

|----------|------------|----------|

#### 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003, Amendment 5

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

| Investigator | Signature | Date |
|---------------------------|-----------|------|
| Printed name: | | |
| Accepted for the Sponsor: | | |

On behalf of BioMarin, I confirm that BioMarin, as a sponsor will comply with all obligations as detailed in all applicable regulations and guidelines. I will ensure that the PI is informed of all relevant information that becomes available during the conduct of this study.

| | | 28 PB 2014 |
|---------------|-----------|------------|
| Medical womon | Signature | Date |
| Printed name: | | |





## 24 PROTOCOL AMENDMENT TEXT REVISIONS

The following table summarizes the revisions made to the protocol and relates the changes to the appropriate rationale (see pages 2-4). Text that has been added or inserted is indicated by <u>underlined font</u>, and deleted text is indicated by <u>strikethrough font</u>.

| Section No./Title | Revision | Rationale |
|---|---|---|
| Global change: Sponsor's Medical Officer | , MD | 16 |
| | This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205. Administration of rAvPAL-PEG will be continued to assess whether long term dosingthe long-term safety and efficacy of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects. | |
| | Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigatorin consultation with the Sponsor's Medical Officer. Diet will be monitored using a diet diary. | |
| Section 2/Symansis Study | A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks-measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001 | |
| Section 2/Synopsis, Study<br>Rationale | | 2, 3, 12 |




This is a long-term extension of rAvPAL-PEG Phase 2 studies in approximately up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies PAL 002 and PAL 004 (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study.

.... The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60 600 µmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL PEG dose for at least 2 consecutive weeks). Doses will be evaluated on an individual basis.

A subject will continue in PAL-003 until one of the following occurs:

- The subject has completed the study through the Month 860 visit.
- The study drug receives marketing authorization.

2, 3, 4, 12

Section 2/Synopsis,

Study Design and Plan

| B <sub>E</sub> OM | ARI | N. |
|-------------------|-----|----|
|-------------------|-----|----|


Subjects who participate in this study will be required to transition into a Phase 3 study (165-302) if weekly doses of rAvPAL-PEG are between 70 mg/week and 350 mg/week (inclusive) provided that doses of rAvPAL-PEG have been stable (ie, no major change in dose for at least 4 weeks). Subjects who meet these criteria must be transitioned from PAL-003 to Study 165-302 provided they meet the 165-302 study eligibility criteria.

<u>Subjects who are eligible for Study 165-302 but do not transition into 165-302 will be withdrawn from this study.</u>

The PAL-003 study will continue until BMN-165 is approved by the Food and Drug Administration (FDA) for marketing in the United States or until the sponsor terminates further development of this drug for the treatment of PKU.

### PAL-003 Substudy

Section 2/Synopsis, Study Design and Plan A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks measurements and for whom no further dose modifications are planned.

2, 3, 4, 12




# **Dose Increase Methodology:**

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Sponsor's Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg) or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg Subjects who increase their dose frequency will have additional assessments performed (Interim Dosing Visit) or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30-60 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.

Section 2/Synopsis, Dose Modifications

2,3,4

| BIOM | ARI | N |
|------|-----|---|
|------|-----|---|

| | Dose Decrease Methodology | |
|---|---|---|
| | All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for safety (ie, hypophenylalanemia or any adverse event that may be improved with a lower, more frequent dose). | |
| | A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration in response to safety, dosing frequency may also be reduced. | |
| Section 2/Synopsis, | If the subject develops low blood Phe (as defined by a blood Phe level $\leq$ 30 $\mu$ mol/Las measured by serum Phe levels for a minimum of 1 month), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician). | |
| Dose Modifications | | 2,3 |
| Section 2/Synopsis,<br>Number of Subjects | | |
| Planned | ApproximatelyUp to 100 subjects. | 17 |




The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self administration: rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver either 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver 15 mg of rAvPAL-PE per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

#### Or

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PE per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

#### Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Section 2/Synopsis, Investigational Product, Dose, Route and Regimen

| Prefilled Syringe | <u>Volume</u> | <b>Concentration</b> | <u>Dose</u> |
|-------------------|---------------|----------------------|--------------|
| <u>Sku #1</u> | <u>0.5 mL</u> | 5 mg/mL | 2.5 mg |
| <u>Sku #2</u> | <u>0.5 mL</u> | 20 mg/mL | <u>10 mg</u> |
| <u>Sku #3</u> | <u>1.0 mL</u> | 20 mg/mL | <u>20 mg</u> |

13

| B:OM/ | ARIN |
|-------|------|
|-------|------|

| Section 2/Synopsis,<br>Investigational Product, | The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection. Upon enrollment into this study, subjects from previous rAvPAL PEG studies will be dosed with the same or higher dose than the dose that was administered upon completion of that study provided that there was no interruption in dosing. Subjects who have had dosing interruptions between the previous rAvPAL PEG study and PAL 003 must have their starting dose determined per the Sponsor's Medical Officer, rAvPAL-PEG doses will be administered SC by either health care professionals or via self administration. The dose level may be increased recreased per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe level (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600 µmol/L for a minimum of 2 weeks consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed byper the PI and the Sponsor's Medical Officer, based upon the subject's response to doses. Fixed Dosing Subjects who have demonstrated efficacy (ie, blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive weeks measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects should convert their weight-based dose using the following table: | |
|---|---|---|
| Regimen | Tabular information regarding fixed doses has been revised. | 3, 13 |
| Section 2/Synopsis,<br>Duration of Treatment | Up to <u>86</u> 60 months. | 1 |


### **Safety Analysis:**

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF). All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of for vital signs, physical examination results, ECG results, and Y-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

# **Efficacy Analysis:**

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the Statistical Analysis Plan [SAP]) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of 60-600 µmol/L will be summarized by each scheduled time point.

# **Exploratory Analysis:**

For subjects who have received any study drug in this study with any post treatment blood Phe concentration measurements and diet diary information, the relationship of dietary Phe intake (per information reported on the subject diet diary), and blood Phe concentration will be explored Details regarding exploratory analyses will be provided in the SAP.

Section 2/Synopsis, Statistical Methods

8, 17

| Section 6, Investigators and Study Administrative Structure | The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Regulatory AffairsPharmacovigilance Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required | 17 |
|---|---|---|
| Section 7.2, Previous | The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002, Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience as of JAN2011 from this ongoing study and the other ongoing Phase 2 studies, PAL-002 and PAL-004. | |
| Clinical Studies | | 17 |
| Section 7.2.2, Phase 2<br>Studies PAL-002,<br>PAL-004, and 165-205 | This section has been updated with results from Studies PAL-002, PAL-004, and PAL 165-205. | 14 |

| BIOM. | ARI | N |
|-------|-----|---|
|-------|-----|---|

| | | T |
|---|---|---|
| | Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also | |
| | on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels | |
| | concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has | |
| | been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe | |
| | level. Changes to subject diet are not allowed in this study unless per the Investigator in consultation | |
| | with the Sponsor's Medical Officer. Diet will be monitored using a diet diary. | |
| | with the sponsor's integreat Officer. Diet will be monitored using a diet diary. | |
| | A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a | |
| | minimum of up to 6 subjects who have achieved and maintained target blood Phe for at least 2 | |
| | consecutive weeks measurements and for whom no further dose modifications are planned. Single- | |
| | dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose | |
| | PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK | |
| | substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe | |
| | reduction to within the protocol-defined target range. | |
| | This study is an extension of previous rAvPAL-PEG Phase 2 studies. Administration of rAvPAL-PEG | |
| | will be continued to assess whether long term dosing the long-term safety and efficacy of | |
| | rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects. | |
| Section 7.3, Study | 1711712 1 20 is sufe and can maintain reduced brood 1 he concentrations in 1 110 subjects. | |
| Rationale | | 2, 3, 12 |
| | Additionally, subjects willmay be premedicated to prevent or mitigate risk of hypersensitivity | |
| Section 7.4.2, Toxicity | reactions (refer to Section 9.1.1.3.3). | |
| Due to an Immunologic | | |
| Reaction | | 10 |

| BIOMARIN <sup>®</sup> PAL-003 A5 Page 112 |
|-------------------------------------------|
|-------------------------------------------|

| Section 7.4.2.2, | Allergic-Hypersensitivity reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or | |
|---|---|---|
| Management of | severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or | |
| Allergic | anaphylaxis. Clinical assessments should be conducted for a minimum of 30-60 minutes post-injection. | |
| <u>Hypersensitivity</u> | | |
| Reactions | | 3, 17 |




This is a long-term extension of rAvPAL-PEG Phase 2 studies in approximately up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies PAL 002 and PAL 004 (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study.

.... The first dose will be administered in the clinic, and the subject must be observed for 30-60 minutes following administration. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator in consultation with the Sponsor's Medical Officer and must be performed under the supervision of the Investigator in consultation with the Sponsor's Medical Officer. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 µmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL PEG dose for at least 2 consecutive weeks). Doses will be evaluated on an individual basis.

A subject will continue in PAL-003 until one of the following occurs:

- The subject has completed the study through the Month 860 visit.
- The study drug receives marketing authorization.

Section 9.1, Overall Study Design and Plan

2, 3, 4, 12

| BIOMARIN | 1º |
|----------|----|
|----------|----|

| | Subjects who participate in this study will be required to transition into a Phase 3 study (165-302) if weekly doses of rAvPAL-PEG are between 70 mg/week and 350 mg/week (inclusive) provided that doses of rAvPAL-PEG have been stable (ie, no major change in dose for at least 4 weeks). Subjects who meet these criteria must be transitioned from PAL-003 to Study 165-302 provided they meet the 165-302 study eligibility criteria. | |
|---|---|---|
| | Subjects who are eligible for Study 165-302 but do not transition into 165-302 will be withdrawn from this study. | |
| | The PAL-003 study will continue until BMN-165 is approved by the Food and Drug Administration (FDA) for marketing in the United States or until the sponsor terminates further development of this drug for the treatment of PKU. | |
| Section 9.1, Overall<br>Study Design and Plan | A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in a minimum of up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive weeks measurements and for whom no further dose modifications are planned | 2, 3, 4, 12 |
| Section 9.1, Table 9.1.1, Schedule of Events | This table has been revised to align with changes made within the amendment. | 15, 17 |
| Section 9.1.1.1, Subjects Who Have Had Previous Hypersensitivity Reactions to rAvPAL-PEG or a PEG-containing | Subjects who had a previous systemic reaction to rAvPAL-PEG or a PEG-containing product that warranted early termination from a previous rAvPAL-PEG study are excluded from participation in this study. Subjects who experienced a generalized skin rash are included in this category. Subjects who have had a previous local skin reaction to rAvPAL-PEG in a previous rAvPAL-PEG study are eligible to participate in this study. | |
| Product | | 17 |

BIOMARIN

PAL-003 A5

| | | 17 |
|---|---|---|
| | All subjects who experience a local skin reaction during this study may be premedicated orally with | 1/ |
| | acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may | |
| | take non-sedating premedications prior to coming to clinic) for all future study doses. Recommended | |
| | premedications are acetaminophen and/or non-sedating antihistamine. The dosage will be standard. | |
| | Subjects must be accompanied by a designated driver (if applicable) b | |
| | cause drowsiness, sedating antihistamines may be administered only if the subject is accompanied by a | |
| | designated driver. Symptoms of local reactions may be treated with local application of ice and | |
| Section 9.1.1.3.1, Local | non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.2.2). | |
| Skin Reactions | | 17 |
| | Subjects will be encouraged to premedicated orally with acetaminophen and/or non-sedating | |
| | antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications | |
| | prior to coming to clinic) for all future study doses. | |
| Section 9.1.1.3.2, Large<br>Local Skin Reactions | | 10 |

| B <b>!</b> OMARIN | PAL-003 A5 | Page 116 |
|-------------------|------------|----------|

Section 9.1.1.3.2.1,
Large Local Skin
Reactions Contiguous
to Injection Site

Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL-PEG or to rAvPAL-PEG or a PEG-containing product may remain in the study if the skin symptoms have resolved and no other symptoms have developed. For the remainder of the study, subjects will be encouraged to premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable).

10

| BIOM | AR | N. |
|------|----|----|
|------|----|----|


....Subjects who experience generalized skin symptoms are included in this category. Immediately after the systemic reaction (within 2448 hours), subjects with generalized skin symptoms must have additional assessments performed for safety (ie, Unscheduled Hypersensitivity Reaction Visit): serum antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG IgE, anti-rAvPAL-PEG neutralizing antibodies); serum tryptase level (it is recommended that this sample be drawn immediately after reaction); sedimentation rate; urine albumin/creatinine ratio; urine N-methyl histamine; CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub>; skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction); and clinical laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1.

.... Subjects who do not have an IgE mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 1 week. If laboratory data shows that the subject experienced an IgE mediated reaction, dosing will not resume until review of the case with the Investigator, Sponsor's Medical Officer, and an allergist/immunologist.

rAvPAL-PEG administration will resume at the next lowest dose level. Restarting of rAvPAL-PEG administration following a systemic reaction must be performed in the clinic for the first week of resumed dosing. Subjects must will be encouraged to premedicated orally with acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30–60 minutes following every administration of study drug. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable).

Section 9.1.1.3.3, Systemic Reactions 4,6,7, 10,

| <b>B</b> OMARIN | PAL-003 A5 | Page 118 |
|-----------------|------------|----------|

| | <del>,</del> | |
|---|---|---|
| | Subjects must will be encouraged to premedicated orally with acetaminophen and/or antihistamines | |
| | 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming | |
| | to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30-60 minutes | |
| | following every study drug administration. Because antihistamines may cause drowsiness, the subject | |
| | must be accompanied by a designated driver (if applicable). | |
| Section 9.1.1.3.3, | | |
| Systemic Reactions | | 4,10 |




## **Dose Increase Methodology:**

Each subject's dose may be modified based on the decision of the Investigator, in agreement with the Sponsor's Medical Officer. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg) or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg Subjects who increase their dose frequency will have additional assessments performed (Interim Dosing Visit) or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30-60 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.

Section 9.1.2.1, Dose Increase Methodology

2,3,4




## Dose Decrease Methodology

All dose decreases must be agreed to by both the Investigator and the Sponsor's Medical Officer. Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for safety (ie, hypophenylalanemia or any adverse event that may be improved with a lower, more frequent dose).

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required to attain the target Phe concentration response to safety, dosing frequency may also be reduced.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/Las measured by serum Phe levels for a minimum of 1 month), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

Section 9.1.2.2, Dose Decrease Methodology

2,3

| BIOMARIN | · · |
|----------|-----|
|----------|-----|


.... The dose level may be increased per Investigator determination in consultation with the Sponsor's Medical Officer based on available information regarding a subject's blood Phe level (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600 µmol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, as agreed to byper the PI and the Sponsor's Medical Officer, based upon the subject's response to doses.

Subjects may self administer study drug at home if approved by the Investigator and the Sponsor's Medical Officer and if adequate training is demonstrated. Subjects may be eligible to self administer study drug if he or she meets the following criteria:

• The subject is on a stable dosing regimen for 2 weeks (ie, the subject has demonstrated a blood Phe level within 60-600 µmol/L for a minimum of 2 consecutive weeks).

Section 9.4, Treatments

3, 5




The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self administration: rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver either 10 mg of rAvPAL-PEG per 1 mL (10 mg/mL protein concentration) or 15 mg or rAvPAL-PEG per 1 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1 mL of the drug product.

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver 15 mg of rAvPAL-PE per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

#### Or

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PE per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

#### Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

| Prefilled Syringe | <u>Volume</u> | Concentration | <u>Dose</u> |
|-------------------|---------------|---------------|--------------|
| <u>Sku #1</u> | <u>0.5 mL</u> | 5 mg/mL | 2.5 mg |
| <u>Sku #2</u> | <u>0.5 mL</u> | 20 mg/mL | <u>10 mg</u> |
| <u>Sku #3</u> | <u>1.0 mL</u> | 20 mg/mL | <u>20 mg</u> |

Section 9.4.2.1, Product Characteristics and Labeling

13

| BIOMARIN | 1º |
|----------|----|
|----------|----|

| | The rAvPAL PEG drug product for SC injection is formulated and supplied as a sterile aqueous | |
|---|---|---|
| | (colorless to pale yellow) solution in clear, single use, type 1 borosilicate glass vials. Each 3 mL vial | |
| | contains 1.5 $\pm$ 0.2 mL to deliver either 10 mg of rAvPAL PEG per 1 mL (10 mg/mL protein | |
| | concentration) or 15 mg of rAvPAL PEG per 1 mL (15 mg/mL protein concentration). Each vial is | |
| | filled with $1.5 \pm 0.2$ mL to allow the withdrawal and delivery of up to 1 mL of the drug product. | |
| Section 9.4.2.1, Product | Dilution instructions are provided in a separate instruction manual. | |
| Characteristics and | | |
| Labeling | | 13 |
| | Doses will be administered SC and the favorable dose will be determined for each subject by adjusting | |
| | the dose level, dose frequency, or both, as agreed by per the PI and the Sponsor's Medical Officer, | |
| | based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg | |
| | (or 375 mg for subjects receiving a fixed dose). | |
| | Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of | |
| | 60-600 µmol/L for at least 2 consecutive weeksmeasurements) and who have maintained a stable | |
| | rAvPAL-PEG dose for at least 2 consecutive weeksmeasurements may be eligible to transition from | |
| | weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). | |
| | Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information | |
| Section 9.4.4, | presented in Table 9.4.4.1. | |
| Directions for<br>Administration | Table 9.4.4.1 has been revised. | 3, 13 |

| BIOMA | ARIN |
|-------|------|
|-------|------|

| | Subjects who have had a prior local skin reaction to rAvPAL-PEG or a PEG-containing product | |
|---|---|---|
| | will be encouraged towill be premedicated with acetaminophen and/or non-sedating antihistamines | |
| | (refer to Section 9.1.1). If the local skin reaction worsens with a repeat injection (as determined by the | |
| | Investigator in consultation with the Sponsor's Medical Officer) even with premedication prior to | |
| | study drug dosing, the subject must be withdrawn from the study and complete an Early Termination | |
| Section 9.4.8, Prior and | Visit. | |
| Concomitant | | |
| Medication | | 10 |
| | During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject | |
| | decision or per the Investigator in consultation with the Sponsor's Medical Officer. Subjects who miss | |
| | more than 2 consecutive weekly doses (weekly dosing schedule) or 3 consecutive daily doses (daily | |
| | dosing schedule) for whatever reason may continue participation in this study. After a dosing | |
| | interruption, rAvPAL-PEG administration should be re-started at the same dose level and dosing | |
| | frequency that was administered prior to the dosing interruption. The first dose of rAvPAL-PEG | |
| | following a dose interruption should be administered in a clinic setting, and the subject must be | |
| | observed for 30-60 minutes following administration due to restarting dosing. A follow-up telephone | |
| | call will be made to the subject to monitor subject safety 24 hours following the return to dosing. | |
| | Subjects should continue to perform the study assessments as outlined in the Schedule of Events (refer | |
| Section 9.4.10, Dose | to Table 9.1.1 during any dosing interruption. | |
| Interruption and Missed | | |
| Doses | | 3, 4 |

| <b>B</b> OMARIN | PAL-003 A5 | Page 125 |
|-----------------|------------|----------|

| Officer | ify subject diet must be made per the Investigator in consultation with the Sponsor's Medical and must be performed under the supervision of the Investigator in consultation with the | |
|---|---|---|
| Section 5.0, Bietary or | or's Medical Officer. | |
| Other Protocol Restrictions | | 3 |
| BIOI | MA | RI | N |
|------|----|----|---|
|------|----|----|---|


Blood samples for Phe concentration measurements will be drawn <u>monthly</u>, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1: ).

Blood Phe may be collected <u>more often than</u> monthly, <u>rather than weekly</u>, at the discretion of the Investigator <del>and provided that the subject meets the following criteria</del> should more frequent monitoring of blood Phe levels be clinically required.

- Is receiving a stable dose of rAvPAL PEG (defined as no dose modifications or interruptions for at least the previous 2 weeks)
- Has a stable blood Phe level (defined as Phe between 60 600 μmol/L for at least 2 consecutive weeks)

The subject may continue to have monthly, rather than weekly, blood Phe collection provided the following do not occur:

- Blood Phe measurement > 600 μmol/L
- Blood Phe measurement ≤ 30 μmol/L

If either of these conditions occurs, then that subject should return to weekly blood Phe draws until the rAvPAL PEG dose has been adjusted and the Phe level is again within the protocol defined target range for at least 2 weeks.

Section 9.7.2.1, Blood Phenylalanine Concentration

| BIOI | MA | RI | N. |
|------|----|----|----|
|------|----|----|----|


| | Immunogenicity will be assessed by determining immune response and neutralizing activity with the | |
|---|---|---|
| | following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG <del>, anti-PAL IgE</del> , anti-PEG IgM, | |
| | anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1.3.3). | |
| | Immunogenicity assays will be performed at the time points indicated in the Schedule of Events | |
| | (Table 9.1.1: ). | |
| Section 9.7.5.2,<br>Antibody Testing | | 7 |
| Section 9.7.6, Clinical | | |
| Laboratory<br>Assessments | Table 9.7.6.1 has been updated to reflect changes made within this amendment. | 6, 17 |
| | The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the | |
| | subject is lost to follow-up, or it has been determined that the study treatment or study participation is | |
| | not the cause of the AE. Resolution Outcome of AEs (and resolution with dates) should be documented | |
| | on the appropriate CRF page(s) and in the subject's medical record <u>unless the subject is lost to follow-</u> | |
| | up or it has been determined that the study treatment or study participation is not the cause of the AE. | |
| Section 10.1, Adverse | | |
| Events | | 9 |

| BIOMARIN |
|----------|
|----------|


| | Pregnancy in a | a subject or partner should be reported within 24 hours of the site becoming aware of the | |
|---|---|---|---|
| | pregnancy to I | BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference | |
| | materials. The | reporting period for pregnancies begins with informed consent and continues until | |
| | 4 weeks follow | wing the last study drug dose. In addition, pregnancy in a subject is also reported on the | |
| | End of Study | CRF. The Investigator must make every effort to follow the subject through resolution of | |
| | _ | (delivery or termination) and to report the resolution to BPV on the Pregnancy Follow- | |
| | | study reference materials. In the event of pregnancy in the partner of a study subject, the | |
| | - | nould make every reasonable attempt to obtain the woman's consent for release of | |
| | | th information. | |
| Section 10.3, | | | |
| Pregnancy | | | 9 |
| | Name: | , MD | |
| | Address: | 105 Digital Drive | |
| | | Novato, CA 94949 USA | |
| | Phone: | | |
| | Fax: | | |
| Section 10.5, BioMarin | E-mail: | | |
| Pharmacovigilance | | | |
| Contact Information | | | 16 |
| | | ister study drug (study drug may be administered on additional days during the week as | |
| | determ | ined by the Investigator, in agreement with the Sponsor's Medical Officer) | |
| Section 12.3.1, Day 1 | | | |
| (Week 1) | | | 3 |


Subjects should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1: The following should be discussed with the subject during the weekly telephone visit:

- Injection-site self inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Confirmation of dose level, frequency, and study drug administration

Weekly visits do not require an in clinic visit if conducted by a home healthcare professional. However, dose modifications must be performed in the clinic. Subjects must have AEs and concomitant medications assessed and an injection site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. For subjects on a stable dose of rAvPAL PEG (ie, no dose change in the last 2 weeks) and have had a phenylalanine (Phe) level at or below target range (60 600 µmol/L) for 2 consecutive weeks—weekly visits may be waived and replaced by a telephone call per discretion of the Investigator but monthly visits are required.

The following study activities will be performed at the weekly visits beginning with Week 2:

- Vital signs
- Injection site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- PK sample

Section 12.3.2, Weekly Telephone Visits

5.15

| BIOMARIN |
|----------|
|----------|


| D: O1 1/ (1 | XIII N | |
|---|---|---|
| | Blood Phe and plasma tyrosine concentration | |
| | <ul> <li>Blood Phe may be collected monthly, rather than weekly, if certain criteria are<br/>satisfied (refer to Section 9.7.2.1).</li> </ul> | |
| | <ul> <li>Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator, in agreement with the Sponsor's Medical Officer)</li> </ul> | |
| | Weekly telephone call | |
| | <ul> <li>For those subjects performing self administration and waiving (per Investigator discretion) the weekly visit (refer to Section 9.1.1.3.3).</li> </ul> | |
| Section 12.3.2, Weekly | | |
| Telephone Visits | | 5, 15 |

| BIOM. | ARI | N |
|-------|-----|---|
|-------|-----|---|


Beginning with Week 4, monthly visits must be performed in the clinic. <u>The following study activities</u> will be performed and consist of all weekly activities listed above in Section 12.3.2 as well as the additional study activities listed below:

- Vital signs
- Injection-site inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration
- PK sample
- Serum anti rAvPAL PEG antibodies (anti PAL IgG, anti PAL IgM, anti PEG IgG, anti PEG IgM, and anti rAvPAL PEG neutralizing antibodies)
- Weekly telephone call

• For those subjects performing self administration and waiving (per Investigator discretion) the weekly visit (refer to Section 12.3.6.

Section 12.3.4, Monthly Visits (Week 4, 8, 12, etc.)

5, 15

| BIOMARIN |
|----------|
|----------|


| | Beginning with Week 12, quarterly visits consist of all weekly (Section 12.3.2) and monthly (Section 12.3.4) activities listed above as well as the additional study activities listed below: | |
|---|---|---|
| | • PK sample | |
| Section 12.3.5, Quarterly Visits (Week | <ul> <li>Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)</li> </ul> | |
| 12, 24, 36, etc) | | 15 |
| Section 12.3.6, Interim Dosing Visit | This visit has been removed | 15 |

| BIOMARIN | B <sub>1</sub> O | M | A | R | N |
|----------|------------------|---|---|---|---|
|----------|------------------|---|---|---|---|


# • Vital signs

- Urine/albumin creatinine ratio
- Sedimentation rate
- Urine N-methyl histamine
- PK sample

Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects who do not have an IgE mediated reaction may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into the clinic for at least 8 weeks. If laboratory data shows that the subject experienced an IgE mediated reaction, dosing will not resume until review of the case with the Investigator, Sponsor's Medical Officer and an allergist/immunologist (refer to Section 9.1.1.3.3).

Section 12.3.7, Unscheduled Hypersensitivity Reaction Visit

6, 15




The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF).

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, physical examination results, ECG results, and X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

Section 14.2, Safety Analysis

| BIOM | ARI | N |
|------|-----|---|
|------|-----|---|


Change in blood Phe concentration from baseline (to be defined in the SAP) to each scheduled time point and presence/absence of antibodies will also be summarized.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis. Information regarding this exploratory analysis will be provided in the Statistical Analysis Plan.

For subjects who completed the Substudy, the effect of stopping and re starting rAvPAL PEG dosing on safety, blood Phe level, and immune response will be explored. Information regarding the analysis Details regarding exploratory analyses will be provided in the SAP Statistical Analysis Plan.

Section 14.4, Efficacy Analysis

| BIOM | ARI | N |
|------|-----|---|
|------|-----|---|


The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study. Meetings of the DMC can be convened at any time at the discretion of the DMC Chair or the Sponsor's Medical Officer. The Chair will be notified by the Sponsor's Medical Officer of all SAEs and will receive summaries of other safety data as available. The DMC will review the study data as soon as it is available during the study, on a schedule defined in the DMC Charter, and offer advice on whether or not to proceed, modify or terminate study enrollment on the basis of toxicity. Details regarding the DMC membership and safety data to be reviewed by members will be provided in a charter.

The responsibilities of the DMC are to:

- Assess the effect and relevance of new external evidence.
- Make recommendations to the BioMarin concerning continuation or termination of the study or other study modifications based on observations.

Section 15, Data Monitoring Committee

| BIOMA | ARIN |
|-------|------|
|-------|------|


| | The treating physician should bill the subject's health insurance company or other third party payer | |
|---|---|---|
| | for the cost of this medical treatment, unless the executed Clinical Trial Agreement between BioMarin | |
| | and the institution of the investigator specifies otherwise. If the subject has followed the Investigator's | |
| | instructions, BioMarin willmay pay for reasonable and necessary medical services to treat the injuries | |
| | caused by the IP or study procedures, if these costs are not covered by health insurance or another third | |
| | party that usually pays these costs. In some jurisdictions, BioMarin is obligated by law to pay for | |
| Section 16, | study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin | |
| Compensation, | will comply with the law. | |
| Insurance, and | | |
| Indemnity | | 17 |
| | BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which | |
| | necessitates access to all original recordings, laboratory reports, and subject records. In addition, all | |
| | source data should be attributable (signed and dated). The Investigator must therefore agree to allow | |
| | direct access to all source data. Subjects (or their legally authorized representative) must also allow | |
| | access to their medical records, and subjects will be informed of this and will confirm their agreement | |
| | when giving informed consent. If an Investigator or institution refuses to allow access to subject | |
| | records because of confidentiality, arrangements must be made to allow an "interview" style of data | |
| Section 17, Case Report | verification. | |
| Forms and Source | | |
| Documents | | 17 |



#### CLINICAL STUDY PROTOCOL

Study Title: Long-term Extension of a Phase 2, Open-Label, Dose-Finding

Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with

PKU

Protocol Number: PAL-003

Investigational Product: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis

phenylalanine ammonia lyase)

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria (PKU)

Sponsor: BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Development Phase: Phase 2

Sponsor's Responsible Medical

Monitor:

, MD

, Clinical Sciences

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Duration: Up to 98 months or until study is terminated

Dose: 0.001 to a maximum weekly dose of 5.0 mg/kg or 375 mg/week

Date of Original Protocol:

October 08, 2008

Date of Amendment 1:

February 09, 2009

Date of Amendment 2:

October 30, 2009

May 04, 2011

Date of Amendment 4:

June 7, 2012

Date of Amendment 5:

February 28, 2014

Date of Amendment 6: Peortuary 28, 2014

October 30, 2014


May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.




# CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Amendment: 6

Date: October 30, 2014

#### RATIONALE AND SUMMARY OF CHANGES

The protocol for Study PAL-003 is being amended to make the following changes:

- 1. All subjects who are on stable doses of rAvPAL-PEG, including subjects on doses between 70 mg/week and 350 mg/week (inclusive) may remain in this study to continue open-label administration with rAvPAL-PEG. Subjects may be eligible for participation in the long-term, open-label extension portion of the Phase 3 study, 165-302. These revisions align with changes being made to the BMN 165 Phase 3 study, 165-302.
- 2. The individual and study stopping criteria have been revised and reflect a better understanding of the risk/benefit with rAvPAL-PEG administration. Stopping criteria revisions are aligned with recommendations from an independent Data Monitoring Committee (DMC) and the Food and Drug Administration (FDA).
  - a. If a severe or life-threatening National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade ≥ 3 hypersensitivity event occurs that is treatment-related and meets clinical criteria (Brown, 2004, J.Allergy Clin.Immunol.) for severe, an ad hoc independent DMC will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct.
  - b. Individual subjects who have an NCI-CTCAE grade ≥ 3 hypersensitivity event that is treatment-related and is suspected to meet the clinical criteria (Brown, 2004, J.Allergy Clin.Immunol.) for severe in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.
  - c. Anaphylaxis (per National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network [NIAID/FAAN] criteria) is an AE of special interest that should be reported to the sponsor within 24 hours to facilitate rapid reporting to sponsor for review.
- 3. Instructions have been added for reintroducing study drug following anaphylaxis.



- 4. Safety precautions have been added:
  - a. Premedications administered prior to study drug for subjects who have had a hypersensitivity AE have been revised based on a better understanding of the safety profile of rAvPAL-PEG. Changes are also consistent with recommendations from an independent immunologist. Should premedication be required, H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) should be administered approximately 2-3 hours prior to study drug per investigator determination. NSAIDs should be given with food and may be omitted if not tolerated.
  - b. At least two epinephrine injectors will be issued to subjects for use in case of anaphylaxis. Subjects will receive training on self-administration and will be instructed to carry one epinephrine injector with them at all times. Sites will assess that the epinephrine injectors have not expired and that subjects are adhering to instructions.
- Information to track and categorize device (prefilled syringe) malfunction and failures, device-related injuries, and any medication errors attributed to device performance has been added.
- 6. Anti-rAvPAL immunoglobulin E (IgE) antibody assessment has been added to the Hypersensitivity Reaction Visit to better assess IgE response. The anti-protein IgE test serves as a control to determine whether anti-rAvPAL IgE antibody positivity may be missed in anti-rAvPAL-PEG IgE assessment due to potential protein epitope masking by the extensive pegylation. The collection and testing of serum anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM and anti-rAvPAL-PEG neutralizing antibodies for Unscheduled Hypersensitivity Visits are no longer necessary as all these antibodies are tested frequently (at routine study visits) and can provide results at or near the time of an hypersensitivity AE.
- 7. rAvPAL-PEG dosing information has been revised to include instructions specific to prefilled syringe. Self-administration training for prefilled syringe drug product has been added.
- 8. The study duration has been extended for another 12 months. The maximum study duration is now 98 months.
- 9. The final follow-up visit schedule has been changed from 1 week to 4 weeks after the final dose to better monitor safety by collecting AEs and SAEs during this period, and to align with the Early Termination Visit as well as other BMN 165 protocols.
- 10. The requirement for observed dosing in clinic following dose interruption has been extended from one day following the interruption to one week following interruption. This revision aligns the requirement for observed dosing following interruption in PAL-003 with that in the 165 phase 3 studies.
- 11. The injection site inspection procedure has been discontinued.



- 12. The criteria for subject eligibility to self-administer study drug has been revised. All subjects in PAL-003 have now been receiving home-based dosing for at least a year; in addition, all subjects in the ongoing Phase 3 BMN 165 studies are dosed at home. Safety data to date indicate that mild to moderate hypersensitivity adverse events commonly occur in subjects receiving BMN 165 but can generally be safely managed with continued home-based dosing. Safety precautions including detailed guidance regarding response to hypersensitivity AEs are being added to all ongoing studies; this guidance supersedes previous PAL-003 instruction mandating return to clinic-based dosing for all hypersensitivity reactions or Grade 3 or higher adverse events. In addition, PAL-003 experience has shown that dosing adjustments (either increase or decrease) are occasionally necessary to maintain optimal Phe control in the long term and can be safely made without return to clinic-based dosing.
- 13. The rAvPAL-PEG immunogenicity profile has been revised and updated. Information that characterizes the specific antibody responses detected in subjects has been added.
- 14. Additional minor changes have been made to improve clarity and consistency.

Specific major revisions since the completion of the last protocol amendment (Amendment 5, dated 28FEB2014) to the text of each section are outlined in Section 24.



#### 2 SYNOPSIS

| NAME OF COMPANY BioMarin Pharmaceutical Inc. | SUMMARY TABLE Referring to Part of the | FOR NATIONAL<br>AUTHORITY USE |
|---|---|---|
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant | Volume:<br>Page:<br>Reference: | |
| Anabaena variabilis phenylalanine ammonia lyase) NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


STUDY SITES: Approximately 20 centers in the United States

PHASE OF DEVELOPMENT: Phase 2

### STUDY RATIONALE:

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data were collected for subjects who have already achieved Phe reduction to within the protocol-defined target range. This substudy has been completed as of 20 December 2013.

|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

### **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

#### STUDY DESIGN AND PLAN:

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study. Subjects' doses will not exceed 375 mg/week.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the sponsor's medical monitor. The first dose will be administered in the clinic, and the subject must be observed for 30 minutes following administration. Additionally, subjects will be given two epinephrine injectors and will be instructed to carry one epinephrine injector with them at all times (refer to Section 9.4). A follow-up telephone call will be made to the

|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self-administration. Additional training will be provided to subjects and demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator or Sponsor.
- The subject has completed the study through the Month 98 visit.

|----------------------------|
|----------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- The study is terminated.
- The study drug receives marketing authorization.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

### PAL -003 Substudy

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed. This substudy has been completed as of 20 December 2013.

### **Dose Modifications:**

#### Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.

|----------------------------|
|----------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first
  modified dose administration. Subjects who increase their dose frequency do not need to be
  observed following injection of study drug if the increase in frequency does not increase the
  overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

# Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600 µmol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be adjusted.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

### Safety Assessment Criteria:

# Response to Hypersensitivity Adverse Events

Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and non-steroidal

|--------------------|
|--------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. NSAIDs should be given with food and may be omitted if not tolerated.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality. Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

# **Individual Stopping Criteria**

Subjects who have an NCI CTCAE grade  $\geq 3$  hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.

### **Dosing in Response to Hypersensitivity Adverse Events**

Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG. Dosing instructions are presented in Table 9.1.1.2.1 and are regardless of previous occurrence.

Once an AE (other than anaphylaxis) improves to grade 1 or resolves, study drug dose may be increased, maintained, or reduced. If dosing has been interrupted due to an AE (other than anaphylaxis) and the investigator determines it is safe for the subject to resume dosing, the first dose after improvement of the AE should be performed in the clinic. The subject must be observed for 30 minutes following administration due to restarting dosing. The subject may be advised to premedicate with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to subsequent BMN 165 doses. NSAIDs should be given with food and may be omitted if not tolerated.

### Response to Anaphylaxis

If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and tryptase (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then be made whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose level.

For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equipment for emergency resuscitation (including epinephrine) within easy access.

|-----------------------------|
|-----------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

The subject must be observed for 30 minutes following administration due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated.

### **Stopping Criteria:**

If an NCI-CTCAE grade ≥3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening or required treatment to prevent a life-threatening event:

- Cyanosis or  $SpO_2 \le 92\%$
- Hypotension with SBP < 90 mm Hg (adults)
- Neurologic alteration: loss of consciousness, collapse, incontinence

Brown's severity criteria are presented in Table 9.1.2.1.

#### NUMBER OF SUBJECTS PLANNED:

Up to 100 subjects.

### DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.
- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of

|-----------------------------|
|-----------------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.

- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the sponsor's medical monitor. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).

|--------------------|
|--------------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG necessitating early termination from a previous rAvPAL-PEG study or known hypersensitivity to any of its excipients.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

### INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self-administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing  $1.5 \pm 0.2$  mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with  $1.5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

### Or:

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PEG per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

#### Or:

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Refer to Table 9.4.2.1.1 for information on prefilled syringe volume, concentration, and dose.

Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be eligible to transition from vial and syringe to prefilled syringe dosing. Additionally, regular refresher training on use of prefilled syringe will be provided in study clinic every 24 weeks, and more often as needed.

| PAL-003 A6 Page 14 | <b>BIOMARIN</b> |
|--------------------|-----------------|
|--------------------|-----------------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

Subjects should convert their vial and syringe dose to prefilled syringe dose using information presented in Table 9.4.2.1.2.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL-PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

#### Fixed Dosing

Subjects who have demonstrated efficacy (ie, blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects should convert their weight-based dose using information presented in Table 9.4.4.1.

#### **DURATION OF TREATMENT:**

Up to 98 months.

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

### **CRITERIA FOR EVALUATION:**

### Efficacy:

Blood Phe concentrations will be measured.

### Immunogenicity:

The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-PEG neutralizing antibodies, anti-rAvPAL IgE, and anti-PEG-PAL IgE) will be assessed.

| BIOMARIN <sup>®</sup> PAL-003 A6 Page 15 | OMARIN' |
|------------------------------------------|---------|
|------------------------------------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

### Safety:

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs, ECG results, X-ray results, and laboratory test results.

### **Pharmacokinetic:**

Plasma concentrations of rAvPAL-PEG will be measured for subjects participating in the Substudy.

### **STATISTICAL METHODS:**

### Sample Size:

Subjects who participated in a previous rAvPAL-PEG study may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

#### **Safety Analysis:**

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by-subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics for vital signs, physical examination results, ECG results, X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

|--------------------|
|--------------------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. | SUMMARY TABLE Referring to Part of the | FOR NATIONAL<br>AUTHORITY USE |
|---|---|---|
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

### **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the Statistical Analysis Plan [SAP]) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

### **Exploratory Analysis:**

Details regarding exploratory analyses will be provided in the SAP.

### **Substudy Analysis:**

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

### **Pharmacokinetic Analysis:**

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F).




# 3 TABLE OF CONTENTS

| 1 | TIT | TLE PAGE | | |
|---|---|---|---|---|
| 2 | SYN | NOPSIS | | |
| 3 | TAF | BLE OF CONTENTS17 | | |
| 4 | LIS | T OF ABBREVIATIONS AND DEFINITIONS OF TERMS21 | | |
| 5 | ETHICS | | | 25 |
| | 5.1 | 5.1 Institutional Review Board or Ethics Committee | | |
| | 5.2 | Ethical | l Conduct of Study | 25 |
| | 5.3 Subject Information and Informed Consent | | | 26 |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 27 |
| 7 | INTRODUCTION | | | 28 |
| | 7.1 | 7.1 Nonclinical Studies | | |
| | 7.2 | Previo | us Clinical Studies | 29 |
| | | 7.2.1 | Phase 1 Study, PAL-001 | 30 |
| | | 7.2.2 | Phase 2 Studies PAL-002, PAL-004, and 165-205 | 30 |
| | 7.3 | Study | Rationale | 34 |
| | 7.4 | 4 Summary of Overall Risks and Benefits | | |
| | | 7.4.1 | Toxicity Due to Exposure to Polyethylene Glycol (PEG) | 35 |
| | | 7.4.2 | Immunologic Response | 36 |
| | | 7.4.3 | Management of Hypersensitivity Reactions | 37 |
| 8 | STU | DY OB | JECTIVES | 39 |
| 9 | INV | ESTIGA | ATIONAL PLAN | 40 |
| | 9.1 Overall Study Design and Plan | | | |
| | | 9.1.1 | Response to Hypersensitivity Adverse Events | 46 |
| | | 9.1.2 | Study Stopping Criteria | 48 |
| | | 9.1.3 | Dose Modifications | 49 |
| | 9.2 | 9.2 Discussion of Study Design, Including Choice of Control Group | | |
| | 9.3 | 9.3 Selection of Study Population | | |
| | | 9.3.1 | Inclusion Criteria | 50 |
| | | 9.3.2 | Exclusion Criteria | 51 |

| В | 0 | MA | RIN | PAL-003 A6 | | Page 18 |
|---|---|---|---|---|---|---|
| | | 9.3.3 | Removal | of Subjects from Treatment of | or Assessment | 52 |
| | | 9.3.4 | Subject Id | entification and Replacemen | nt of Subjects | 53 |
| | 9.4 | Treatme | ents | | | 53 |
| | | 9.4.1 | Treatment | s Administered | | 55 |
| | | 9.4.2 | Identity of | f Investigational Product (IP) | ) | 55 |
| | | 9.4.3 | Storage | | | 58 |
| | | 9.4.4 | Directions | for Administration | | 58 |
| | | 9.4.5 | Method of | f Assigning Subjects to Treat | tment Groups | 59 |
| | | 9.4.6 | Selection | of Doses Used in the Study . | | 60 |
| | | 9.4.7 | Blinding | | | 60 |
| | | 9.4.8 | Prior and | Concomitant Medications | | 60 |
| | | 9.4.9 | Treatment | Compliance | | 61 |
| | | 9.4.10 | Dose Inter | rruption and Missed Doses | | 61 |
| | 9.5 | Investig | gational Pro | duct Accountability | | 61 |
| | | 9.5.1 | Return and | d Disposition of Clinical Sup | oplies | 62 |
| | 9.6 | Dietary | or Other P | rotocol Restrictions | | 62 |
| | 9.7 | Efficac | y and Safet | y Variables | | 62 |
| | | 9.7.1 | Efficacy a | nd Safety Measurements Ass | sessed | 62 |
| | | 9.7.2 | Efficacy V | <sup>7</sup> ariable | | 64 |
| | | 9.7.3 | Pharmaco | kinetic Variables | | 64 |
| | | 9.7.4 | Explorator | ry Efficacy Variable | | 64 |
| | | 9.7.5 | Safety Va | riables | | 65 |
| | | 9.7.6 | Clinical L | aboratory Assessments | | 65 |
| 10 | REP | ORTING | G ADVERS | SE EVENTS | | 67 |
| | 10.1 | Adverse | e Events | | | 67 |
| | 10.2 | Serious | Adverse E | vents | | 69 |
| | 10.3 | Pregnar | ncy | | | 71 |
| | 10.4 | Urgent | Safety Mea | sures | | 71 |
| | 10.5 | BioMar | in Pharmac | covigilance Contact Informat | tion | 72 |
| 11 | APP | ROPRIA | TENESS ( | OF MEASUREMENTS | | 73 |

| B | OMARIN | PAL-003 A6 | Page 19 |
|---|---|---|---|
| | 11.1 Safety and Pharm | acokinetics | 73 |
| | - | | |
| 12 | _ | ES | |
| | 12.2 Screening Visit | | 74 |
| | _ | | |
| | 12.3.1 Day 1 (W | <sup>7</sup> eek 1) | 75 |
| | 12.3.2 Weekly 7 | Felephone Visit | 75 |
| | 12.3.3 Substudy | Visits | 76 |
| | 12.3.4 Monthly | Visits (Week 4, 8, 12, etc) | 76 |
| | 12.3.5 Quarterly | Visits (Week 12, 24, 36, etc) | 76 |
| | 12.3.6 Unschedu | aled Hypersensitivity Reaction Visit | 77 |
| | 12.4 Early Termination | ı Visit | 77 |
| | 12.5 Final Follow-up V | /isit | 78 |
| 13 | DATA QUALITY ASS | SURANCE | 80 |
| 14 | STATISTICAL METH | ODS AND DETERMINATION OF SA | MPLE SIZE81 |
| | 14.1 Statistical and An | alytical Plans | 81 |
| | 14.2 Safety Analysis | | 81 |
| | 14.3 Pharmacokinetic | Analysis | 81 |
| | 14.3.1 Pharmace | okinetic Substudy Analysis | 82 |
| | 14.4 Efficacy Analysis | | 82 |
| | 14.5 Determination of | Sample Size | 82 |
| | 14.6 Handling of Miss | ing Data | 82 |
| | 14.7 Interim Analyses | | 83 |
| | 14.8 Changes in the Co | onduct of the Study or Planned Analyses | 83 |
| 15 | DATA MONITORING | COMMITTEE (DMC) | 84 |
| 16 | COMPENSATION, IN | SURANCE, AND INDEMNITY | 85 |
| 17 | CASE REPORT FORM | AS AND SOURCE DOCUMENTS | 86 |
| 18 | STUDY MONITORIN | G AND AUDITING | 87 |
| 19 | RETENTION OF REC | ORDS | 88 |

|---|---|---|
| 20 USE OF INFORMATION | ON AND PUBLICATION | 89 |
| 21 REFERENCES | | 90 |
| 22 INVESTIGATOR RESI | PONSIBILITIES | 92 |
| 22.1 Conduct of Study | and Protection of Human Subjects | 92 |
| 24 PROTOCOL AMENDA | MENT MAJOR TEXT REVISIONS | 94 |
| LIST OF TABLES | | |
| Table 9.1.1: Schedule of Ev | vents | 42 |
| Table 9.1.2: PK Substudy I | Oosing Regimens | 45 |
| Table 9.1.1.2.1: Dosing Ins | tructions in Response to Hypersensitiv | vity Adverse Events47 |
| Table 9.1.2.1: Brown's Sev | verity Criteria | 49 |
| Table 9.4.2.1.1: Prefilled S | yringe Volume, Concentration, and Do | ose56 |
| Table 9.4.2.1.2: Conversion | n from Vial and Syringe Dose to Prefil | led Syringe Dose56 |
| Table 9.4.4.1: Fixed Doses | for Subjects on Weight-Based Dose R | egimen59 |
| Table 9.7.1.1: Summary of | Laboratory Assessments | 63 |
| Table 9.7.6.1: Clinical Lab | oratory Tests | 66 |




### 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase

AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

 $AUC_{0-7 \text{ days}}$  area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen

°C degree Celsius

C<sub>3</sub> complement 3

C<sub>4</sub> complement 4

CBC complete blood count

CD Compact disk

CFR Code of Federal Regulations

CH50 total hemolytic complement

C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form

CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure




DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up

g gram

GCP Good Clinical Practice

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure

ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

ID identification

IgE immunoglobulin E

IgG immunoglobulin G

IgM immunoglobulin M

IP investigational product

IRB Institutional Review Board

IV intravenous

kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

NAb neutralizing antibodies





NCI National Cancer Institute

NIAID/FAAN National Institute of Allergy and Infectious Disease/Food Allergy and

Anaphylaxis Network

NOAEL no observable adverse effect level

NSAID non-steroidal anti-inflammatory medication

OTC over the counter

PAH phenylalanine hydroxylase

PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator

PK pharmacokinetics

PKU phenylketonuria

rAvPAL-PEG recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG

RBC red blood cell

SAE serious adverse event

SAP Statistical Analysis Plan

SBP systolic blood pressure

SC subcutaneous

SD standard deviation

SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase

SGPT serum glutamic pyruvate transaminase

US United States

WBC white blood cell



# **Definition of Terms:**

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.


#### 5 ETHICS

# 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

# 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will



provide written, informed consent before any study-related tests or evaluations are performed.

## 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR Part 50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



#### 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Pharmacovigilance Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations and urinalysis. Pharmacokinetic (PK) analysis will be performed by BioMarin.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.



#### 7 INTRODUCTION

A comprehensive review of PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

### 7.1 Nonclinical Studies

The nonclinical program for rAvPAL-PEG has characterized the pharmacology, pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC route of administration. Pharmacology was assessed in the BTBR *Pah*<sup>enu2</sup> (ENU2) mouse model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to 2000 μΜ) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to male ENU2 mice, plasma Phe concentrations decreased from approximately 2000 μΜ to < 200 μΜ after 2 dose administrations. An attenuated reduction of blood Phe was seen between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe < 200 μM over the entire week, which continued for a total of 15 weeks.

In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a 2-4 week dose interruption and an 11-week dose interruption. Following both dose interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A similar interim attenuated response was observed with the longer dose interruption of approximately 11 weeks. In both of these assessments, no safety issues were noted upon re-starting dosing with rAvPAL-PEG (Lapis, 2007, ASHG 57th Annual Meeting).

Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No respiratory or central nervous system (CNS) effects were seen with SC administration of rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV effects of rAvPAL-PEG administered subcutaneously.

Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats and cynomolgus monkeys. The elimination half-life ( $t_{1/2}$ ) values of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and 44 hours, respectively,

and exhibited modest area under the plasma concentration-time curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the  $t_{1/2}$  was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum observed plasma concentration ( $C_{max}$ ), along with a long  $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) the AUC and the  $C_{max}$  are roughly linearly proportional.

Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given ≥ 3 mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey.

#### 7.2 Previous Clinical Studies

The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan<sup>®</sup> or are not compliant with Kuvan<sup>®</sup> treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002, Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience from this ongoing study and the other ongoing Phase 2 studies, PAL-002 and PAL-004.



### 7.2.1 Phase 1 Study, PAL-001

The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations.

The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 µmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG.

Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows:

- rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg.
- For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level for these 5 subjects was 1113 μmol/L.
- Overall, no clinically significant reductions in blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, 0.01, and 0.03 mg/kg.
- For subjects who were administered rAvPAL-PEG at the 3 higher dose levels (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration levels, the calculated PK parameters were a mean T<sub>max</sub> of 89-106 hours, a t<sub>1/2</sub> of 46-120 hours, and an AUC<sub>0-t</sub>, and C<sub>max</sub> that were proportional with dose. Drug exposure was slightly increased with increased dose.

#### 7.2.2 Phase 2 Studies PAL-002, PAL-004, and 165-205

Based on results from the Phase 1, single-dose study, the Phase 2 studies have been designed to evaluate rAvPAL-PEG at various doses and dosing regimens to safely achieve and maintain blood Phe reductions in subjects with PKU. Currently, there are three ongoing Phase 2 studies (PAL-002, PAL-004, 165-205); an overview of each study is presented in Section 7.2.2.1 (PAL-002), Section 7.2.2.2 (PAL-004), and Section 7.2.2.3 (165-205).



### 7.2.2.1 Study PAL-002

Study PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria) was initiated in September 2009 and has completed enrollment. As of 10 September 2012, 40 subjects have been enrolled and 37 have completed the study. PAL-002 enrolled 11 previously exposed subjects from the single-dose study, PAL-001, and 29 subjects who were naïve to rAvPAL-PEG. Thirty-three of the 37 subjects who completed PAL-002 enrolled into this open-label extension study (PAL-003). Two subjects discontinued from the study due to lost to follow-up, relocation, or other reasons, and 1 subject discontinued from the study due to an AE (skin reaction).

The primary objective of this study was to evaluate the effect of multiple doses of rAvPAL-PEG (ranging from 0.001 mg/kg/week to 1.0 mg/kg/week) on blood Phe concentrations in subjects with PKU with up to 16 weeks of treatment. The secondary objectives of the study were to evaluate the safety and tolerability of SC injections of multiple doses of rAvPAL-PEG, to evaluate the immune response to rAvPAL-PEG, and to evaluate the PK profile of rAvPAL-PEG in subjects with PKU.

The PAL-002 study design consists of two parts. In Part 1, rAvPAL-PEG was administered as a once weekly fixed, low-dose induction regimen for 8 weeks. In Part 2, the rAvPAL-PEG dose was titrated upwards; subjects received adjustable dose increases for up to 8 weeks to achieve a target blood Phe concentration of 600 µmol/L. The doses and dosing schedules were revised with a series of protocol amendments to incorporate the information gained during conduct of this early, open-label, multiple-dose study.

A wide range of doses was planned for the PAL-002 study, beginning with doses as low as  $0.001 \, \text{mg/kg/week}$ . However, no substantial reductions in blood Phe level were observed in the majority of subjects who were administered rAvPAL-PEG in the initial four cohorts at doses of 0.001, 0.003, 0.01, and 0.03 mg/kg administered once per week. The absence of appreciable Phe reduction after 16 weeks of treatment in this range of doses led to a decision to amend the study protocol to include a cohort with a higher starting dose of  $0.1 \, \text{mg/kg/week}$ , which had been previously shown to decrease blood Phe levels to approximately  $600 \, \mu \text{mol/L}$  in the single-dose, Phase 1 study (PAL-001). After the first 2 weeks of dosing at  $0.1 \, \text{mg/kg/week}$ , transient Phe reduction was observed in this subset of subjects. However, this dosing regimen was accompanied by mild to moderate hypersensitivity reactions primarily after the second weekly dose, suggesting that additional exploration of dosing regimens would be required.

PAL-003 A6


In summary, preliminary results from PAL-002 demonstrated that doses below 0.1 g/kg administered once per week were not effective in reducing Phe levels. While transient reduction of Phe was apparent at doses of at least 0.1 mg/kg given once per week, this dose regimen was associated with a high incidence of systemic hypersensitivity reactions, typically following the second weekly dose. Further escalation above this dose of 0.1 mg/kg/week would be required to sustain the effect on Phe levels over time. Increased doses would require spreading dose administration over several days per week, as once-weekly administration of higher doses would not be practical due to the large volume of study drug. Therefore, additional dosing regimens would need to be explored in a subsequent study (PAL-004).

Once subjects completed Study PAL-002, they were eligible to enroll into this open-label extension study, PAL-003 to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

## 7.2.2.2 Study PAL-004

PAL-004 (An Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Dose Levels of rAvPAL-PEG Administered Daily in Subjects With Phenylketonuria) was initiated in April 2011 and has completed enrollment. As of 10 September 2012, 16 subjects have been enrolled, 15 subjects have completed the study, and 15 subjects have enrolled into this study (PAL-003). One subject withdrew consent from continued participation prior to study completion. All subjects enrolled in this study were naïve to rAvPAL-PEG exposure.

The objective of this study was to determine if daily administration (defined as 5days/week) of rAvPAL-PEG at dose levels of 0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day was safe and effective in reducing and maintaining blood Phe concentrations to 600 µmol/L in subjects with PKU. The starting dose was 0.4 mg/kg, administered 5 days/week. A total of 12 subjects were added in sequence and were started on doses of 0.4, 0.2, 0.1, 0.06 mg, or 0.001/kg/day based on incoming safety data. Overall, subjects in PAL-004 who initiated treatment at higher daily doses of 0.1 to 0.4 mg/kg/day achieved immediate and substantial reduction of blood Phe levels, but dosing had to be temporarily reduced or interrupted due to the onset of systemic hypersensitivity reactions at approximately Day 10 of dosing. Phe reductions did not persist in the setting of temporary dose reduction or interruption, but Phe levels generally improved if higher dose levels were reinstated.

To prevent the onset of hypersensitivity reactions that were temporally associated with the onset of anti-drug IgM responses, an additional dosing strategy was assessed in PAL-004;



PAL-003 A6


4 subjects initiated dosing at a low dose of 0.001mg/kg/day or 0.06mg/kg/day for 5 consecutive days and then dosing was suspended for 2 weeks. Dosing was restarted on Day 21 at the initial dose followed by dose titration to target Phe levels. Subjects administered this dosing regimen had similar efficacy, but the incidence of hypersensitivity reactions appeared to be similar to that of subjects who did not have the planned dose interruption, suggesting little advantage with this alternate induction regimen.

Experience from PAL-004 indicated that initiating daily rAvPAL-PEG dosing with relatively high daily doses was not sustainable due to the onset of hypersensitivity reactions that occurred approximately 9 to 12 days after the start of administration, nor was the alternate dosing regimen (2 week drug holiday) well tolerated or effective in Phe reduction. In addition, the daily treatment regimen did not reduce the time to achieve target blood Phe levels seen in previous studies. This study indicated that to improve tolerability, rAvPAL-PEG should be initiated with an induction period at doses substantially lower than 0.4mg/kg, followed by upward dose titration toward target Phe levels.

Once subjects completed Study PAL-004, they were eligible to enroll into this open-label extension study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

# 7.2.2.3 Study 165-205

Study BMN 165-205 (A Phase 2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate Safety, Efficacy, and Tolerability of Subcutaneously Administered rAvPAL-PEG in Subjects With PKU for 24 Weeks) was initiated in May 2012. Data from ongoing Studies PAL-002, PAL-004, and PAL-003 suggested that a 4-week treatment course with weekly dosing at a fixed low dose (induction), followed by a weekly 2-fold, upward titration of rAvPAL-PEG to approximately 10-fold higher than the initiation dose (maximum of 375 mg/week) is effective and well tolerated. The objective of this study was to further assess this dosing regimen. Two rAvPAL-PEG dosing regimens were to be explored in this study: weekly low-dose induction (2.5 mg/week for 4 to 8 weeks), followed by a period of upward dose titration towards a target Phe level (600 µmol/L) followed by maintenance dosing at that level through the 24 week study duration (Group 1). The other dosing regimen planned for this study (Group 2) involved administration of a single bolus dose of 8 mg, followed by a treatment holiday of at least 3 weeks duration followed by resumption and escalation of study drug administration following a pattern similar to that employed in Group 1. A total of 24 subjects were enrolled into 165-205. In addition to confirming an effective, well-tolerated dose regimen, this study incorporated non-weight-based dosing, starting with dose



administration once per week at a low dose (2.5mg) with gradual escalation and conversion of dose administration to 5x/week dosing for chronic maintenance therapy.

Once subjects have completed Study 165-205, they are eligible to enroll into this study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week, or into the Phase 3 study, BMN 165-302.

# 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH. Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan<sup>®</sup> is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. rAvPAL-PEG is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an 



exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

This study is an extension of previous rAvPAL-PEG Phase 2 studies. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

# 7.4 Summary of Overall Risks and Benefits

It is not expected that data from previous rAvPAL-PEG studies will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

### 7.4.1 Toxicity Due to Exposure to Polyethylene Glycol (PEG)

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg rAvPAL-PEG SC. In rats, both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1).



In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

## 7.4.2 Immunologic Response

The active drug substance in rAvPAL-PEG is a bacterial protein and elicits immune recognition and subsequent antibody responses. Antibody epitopes on the protein are expected to be rendered at least partially inaccessible by the extensive PEGylation on the drug (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model but does not eliminate antibody formation. Although PEGylation of rAvPAL likely reduces the antigenicity of the molecule, 100% of individuals exposed to rAvPAL-PEG develop antibodies against rAvPAL.

Drug-specific immune responses can range from clinical irrelevance to causing serious hypersensitivity AEs (such as anaphylaxis) and may reduce efficacy due to antibody-mediated drug clearance or antibody neutralization of enzymatic activity. Historically, PEG was thought to be nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.), (Harris, 2003, Nat.Rev.Drug Discov.); however, repeated studies have found that subcutaneous (SC) and intravenous exposure to PEG can induce anti-PEG antibodies (Harris, 2003, Nat.Rev.Drug Discov.), (Richter, 1983, Int.Arch.Allergy Appl.Immunol.). In some instances, development of such antibodies did not result in significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). However, PEG antibody responses were associated with hypersensitivity reactions to PEGylated liposomes (Judge, 2006, Mol.Ther.). Anti-PEG antibodies have also been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.).

Subjects participating in the Phase 2 clinical studies have been monitored closely for anti-drug immunogenicity (anti-rAvPAL immunoglobulin G [IgG], anti-rAvPAL IgM, anti-PEG IgM, anti-PEG IgG, neutralizing antibodies that inhibit PAL enzymatic activity, anti-rAvPAL IgE, and anti-rAvPAL-PEG IgE), complements, C-reactive protein (CRP), ESR, and complete chemistry. All subjects treated with rAvPAL-PEG in the Phase 2 clinical trials developed antibodies against the PAL protein. Anti-rAvPAL IgM antibodies were first detected within 2-3 weeks of treatment initiation and anti-rAvPAL IgG antibodies were detected within 2-3 months. The anti-rAvPAL IgG response generally peaked by 3-5 months and was sustained in all subjects. Neutralizing antibodies (NAb) capable of inhibiting enzymatic activity were detected in a minority of subjects 2-3 months after treatment

|----------|------------|---------|
|----------|------------|---------|

initiation. The timing of the NAb response suggests these antibodies may be a component of the anti-rAvPAL IgG response. It is expected that the centralized location of the PAL active site, within the tetrameric structure, makes it difficult for antibodies to bind and inhibit enzymatic activity. In addition, anti-PAL antibody binding is likely sterically hindered by the extensive PEGylation. The majority of treated subjects also developed a transient anti-PEG antibody response. The anti-PEG response was comprised of IgM and IgG isotypes. In general, anti-PEG antibodies were no longer detected after 5-6 months of treatment. This type of transient antibody response is typical of T cell-independent type 2 (TI-2) responses.

The majority of immune-mediated AEs experienced in subjects treated with rAvPAL-PEG in the Phase 2 studies are believed to be the result of antibody-mediated hypersensitivity. The primary immune mediator is thought to be IgM immune complexes, as evidenced by the timing of onset prior to IgG development and the reduced occurrence over time. IgE positive test results have not been associated with hypersensitivity in any of the subjects thus far, and the majority of subjects have been safely rechallenged with rAvPAL-PEG following reactions. IgM immune complexes are known to be efficient activators of the classical complement pathway and can lead to the accumulation of complement component anaphylatoxins (C3a, C4a, C5a) that can induce hypersensitivity symptoms. Although IgG immune complexes can also activate the classical complement pathway, they do so with less efficiency than IgM. This is due, in part, to the requirement for multiple Fc regions in close proximity to activate the complement cascade, meaning that multiple monomeric IgG Abs are required to bind, whereas only one pentameric IgM Ab is needed to bind to activate complement. Also, in the case of rAvPAL-PEG, binding of anti-PAL IgG antibodies is likely compromised due to epitope masking by the PEGylation, which may reduce IgG-mediated complement activation in vivo. This complex dynamic between combined isotype-specific Ab responses and epitope accessibility is thought to be a major factor dictating the need for an induction and titration dose regimen in the treatment of rAvPAL-PEG to be implemented in this study.

### 7.4.3 Management of Hypersensitivity Reactions

Hypersensitivity reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 30 minutes post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of hypersensitivity reactions. Because of the potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and 



PAL-003 A6


after the rAvPAL-PEG injection. Subject should be pre-medicated with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated. Subjects who qualify for self-administration of study drug are trained to recognize a serious hypersensitivity AEs and how to respond. Additionally, subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (Section 9.4). Refer to Section 9.1.1.3 for instructions regarding resumption of study drug following resolution of symptoms consistent with a clinical diagnosis of anaphylaxis per National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria (Sampson, 2006, J.Allergy Clin.Immunol.).

In the event of a hypersensitivity reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for immunology studies and complement testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of hypersensitivity reaction symptoms:

- Maintain the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oral or IV glucocorticoids.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. An allergy and/or immunology consultation should be sought if necessary. Detailed instructions for the management of hypersensitivity reactions are provided in the Study Reference Manual.



#### 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objective is as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.



#### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity was observed in a previous rAvPAL-PEG studies. Subjects' doses will not exceed 375 mg/week.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the sponsor's medical monitor. The first week of dosing will be administered in the clinic, and the subject must be observed for 30 minutes following administration. Subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (refer to Section 9.4). A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to clinic monthly for review with the clinical study staff.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self-administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self-administration. Additional information is provided in the Subject Self-Administration Training Materials. Additional training will be provided and demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.



In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 9.1.1 and Table 9.1.2. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator or Sponsor.
- The subject has completed the study through the Month 98 visit.
- The study is terminated.
- The study drug receives marketing authorization.

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed (refer to Table 9.1.2).

The Schedule of Events and PK substudy collection schedules are presented below in Table 9.1.1 and Table 9.1.2

PAL-003 A6


**Table 9.1.1: Schedule of Events** 

| | | | | Treatment Pe | eriod <sup>b,c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Monthly b<br>(eg, Wk 4,<br>8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Interim<br>Clinician<br>Visit (HHRN<br>or Site) | Final F/U<br>Visit | Self-<br>administration | Early<br>Term.<br>Visit | Unsched. |
| Assessments and Events | Screening <sup>a</sup> | D 1 | Starting at<br>Week 2 | Every 4th week; | Every 12th week. Perform in addition to monthly procedures | Up to daily | 4 weeks<br>after final<br>dose | | 4 weeks<br>after<br>final<br>dose | Hyper.<br>Reaction<br>Visit. <sup>d</sup><br>Perform<br>within<br>24 hours |
| Informed consent | X | | | | | | | | | |
| Medical history, including | | | | | | | | | | |
| allergy history, and | X | | | | | | | | | |
| demographics | | | | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | | X | | X | | X | |
| Vital signs <sup>e</sup> | X | X | | X | | X | | | X | X |
| Weight | X | | | X | | | | | | |
| 12-lead ECG | X | | | | | | X | | X | |
| Clinical laboratory tests <sup>f</sup> | X | | | X | | | X | | X | $X^{g}$ |
| Complements C <sub>3</sub> and C <sub>4</sub> <sup>h</sup> | X | | | | X | | | | | $X^g$ |
| Sedimentation rate | | X | | | X | | X | | X | |
| Chest x-ray | X | | | X<br>(Week 48<br>visit only) | | | X | | X | |
| Urine pregnancy test <sup>i</sup> | X | X | | X | | | X | | X | |
| Adverse events <sup>j,k</sup> | X | X | X | X | | X | X | X | X | X |
| Weekly phone call to self | | | | | | | | | | |
| admin participants only (to assess AEs, Inj site reactions, | | | X | | | | | X | X | |
| concomitant medications) | | | | | | | | | | |
| Concomitant medications | X | X | X | X | | X | X | X | X | X |
| Diet query | X | X | | X | | | X | | X | |

BIOMARIN

PAL-003 A6


| | I | 1 | | Treatment Pe | | | 1 | | <u> </u> | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Monthly b (eg, Wk 4, 8, etc.) | Quarterly (eg, Wk 12, 24, etc.) Every 12th | Interim<br>Clinician<br>Visit (HHRN<br>or Site) | Final F/U<br>Visit | Self-<br>administration | Early<br>Term.<br>Visit | Unsched.<br>Hyper. |
| Assessments and Events | Screening <sup>a</sup> | D1 | Starting at<br>Week 2 | Every 4th<br>week; | week. Perform in addition to monthly procedures | Up to daily | 4 weeks<br>after final<br>dose | | 4 weeks<br>after<br>final<br>dose | Reaction Visit. <sup>d</sup> Perform within 24 hours |
| 3-Day diet diary <sup>l</sup> | | | | X | | • | X | | X | |
| Serum antibodies <sup>m</sup> | | X | | | X | | X | | X | X |
| Plasma Phe and plasma tyrosine <sup>n</sup> | X | X | | $X^{m}$ | | | X | | X | |
| Urine albumin/creatinine ratio | | | | | | | | | | X |
| Urine N-methyl histamine | | | | | | | | | | X |
| Plasma PK sample <sup>o</sup> | | X | | | X | | X | | X | |
| Administer study drug <sup>p</sup> | | X | | X | | X | | X | | |
| Training (prefilled syringe) <sup>q</sup> | | | | X<br>Transition to<br>prefilled<br>syringe | X<br>Every 24<br>weeks only | | | | | |
| Skin biopsy (optional; affected and not affected area) | | | | | | | | | | X |
| Serum tryptase level <sup>r</sup> | | _ | | | | | | | | X |

AE, adverse event; C<sub>3</sub>, complement 3; C<sub>4</sub>, complement 4; CH50, total hemolytic complement; CRP, C-reactive protein; D, day; ECG, electrocardiogram; ETV, Early Termination Visit; F/U, Follow-up; Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> A separate Screening visit for this study is required only if the time between completion of the previous rAvPAL-PEG study and enrollment into PAL-003 is greater than 28 days.

<sup>&</sup>lt;sup>b</sup> Monthly visits must be performed in the clinic.

| BIOMARIN' PAL-003 A6 Page 44 |
|------------------------------|
|------------------------------|

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

- <sup>g</sup> Subjects who have a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade ≥ 3 hypersensitivity AE should be assessed for CRP, CH50, C1, C3, and C4 within 24 hours of the reaction.
- <sup>h</sup> Complement C3 and C4 will be collected at the Screening Visit and quarterly. Additional complement testing will be performed and as needed to resolve previous abnormal test results.
- <sup>i</sup> If positive or equivocal, perform serum pregnancy test.
- <sup>j</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm).
- <sup>k</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or the final study visit. The reporting period for nonserious AEs is from the first administration of study drug through 4 weeks after last dose or the early termination visit. The reporting period for device-related events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe.
- <sup>1</sup> It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.
- <sup>m</sup> For unscheduled hypersensitivity reaction visit, draw serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only; sampling must be performed > 8 hours after event onset and before the next dose of study drug.
- <sup>n</sup> Samples should be drawn at least 2.5 hours after a meal. At the Investigator's discretion, blood Phe may be collected more often should more frequent monitoring of blood Phe levels be clinically warranted.
- ° Sampling should be performed predose.
- <sup>p</sup> Dosing is up to 5.0 mg/kg/week or 375 mg/week, including subjects who receive more than 1 dose/week. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may be re-evaluated.
- <sup>q</sup> Initial training on the use of prefilled syringe occurs at the next monthly visit and each subsequent day after transition until (in clinic or by HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter.
- <sup>r</sup> Mandatory for subjects who have a hypersensitivity AE. Perform within 24 hours of event onset.

<sup>&</sup>lt;sup>d</sup> Refer to Section 9.1.1 and Section 12.3.6.

<sup>&</sup>lt;sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.

<sup>&</sup>lt;sup>f</sup> Clinical laboratory tests to include spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis. Urine microscopy will be performed if any urinalysis results are positive for hematuria. Refer to Table 9.7.6.1.



PAL-003 A6


**Table 9.1.2: PK Substudy Dosing Regimens** 

| <b>Treatment Frequency</b> | Plasma PK Sampling | Example |
|---|---|---|
| Subjects who are administered study drug once per week | Pre-dose and every 24 hours<br>thereafter (24, 48, 72, and 96<br>hours when possible), and pre-<br>dose of the next weekly dose | If dosed on Monday: Obtain PK sample pre-dose when possible – pre-dose Monday, Tuesday, Wednesday, Thursday, Friday, and pre-dose the following Monday. No further PK substudy draws. |
| Subjects who are<br>administered study drug<br>two or three times per<br>week | Pre-dose and every 24 hours during the longest period between doses, when possible, and pre-dose of the next dose. | If dosed on Monday, Thursday, and Friday: Obtain PK sample every 24 hours during the longest period between doses: Predose Monday, Tuesday, Wednesday, and pre-dose Thursday. No further PK substudy draws. |
| Subjects who are administered study drug four to seven times per week. | Pre-dose and every 12 hours during the longest period between doses, when possible, then pre-dose of the next dose. | If dosed Monday through Friday: Obtain PK sample every 12 hours during the longest period between doses (Friday to Monday): pre-dose Friday, 12 hours post-dose Friday, Saturday (24 and 36 hours post dose), Sunday (48 and 60 hours post-dose), and pre-dose the following Monday. No further PK substudy draws. |



### 9.1.1 Response to Hypersensitivity Adverse Events

Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. NSAIDs should be given with food and may be omitted if not tolerated.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality (Section 9.1.1.3). Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

# 9.1.1.1 Individual Stopping Criteria

Subjects who have an NCI CTCAE grade  $\geq 3$  hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.

#### 9.1.1.2 Dosing in Response to Hypersensitivity Adverse Events

Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG. Dosing instructions are presented in Table 9.1.1.2.1 and are regardless of previous occurrence:

|-----------------------------|
|-----------------------------|

Table 9.1.1.2.1: Dosing Instructions in Response to Hypersensitivity Adverse Events

| | | Action | with Study | Drug | | |
|---|---|---|---|---|---|---|
| NCI-<br>CTCAE<br>Grade <sup>a</sup> | Related to<br>Study Drug | Maintain <sup>b</sup> | Reduce <sup>c</sup> | Interrupt <sup>c</sup> | Individual<br>Stopping<br>Criteria <sup>d</sup> | HRV Assessment <sup>e</sup> |
| 1 | Yes or No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 2 | Yes or No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 3 | No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 3 | Yes | X | (X)<br>Optional | (X)<br>Optional | | Yes |
| and is<br>suspected to<br>meet<br>Brown's<br>criteria for<br>severe | Yes | | | | X<br>Consult with<br>sponsor<br>medical<br>monitor | Yes |
| 4 <sup>d</sup> | Yes or No | | | | X<br>Consult with<br>sponsor<br>medical<br>monitor | Yes |

AE, adverse event; CTCAE, Common Terminology Criteria for Adverse Events, version 4.03; HRV, Hypersensitivity Reaction Visit; NCI, National Cancer Institute.

<sup>&</sup>lt;sup>a</sup>NCI-CTCAE grade determination is performed by the investigator and may be done either via telephone or clinic visit.

<sup>&</sup>lt;sup>b</sup>The investigator will instruct the subject to maintain the rAvPAL-PEG dose at the time of AE onset until improvement to grade 1 or resolution (per investigator assessment in the clinic or via telephone).

<sup>&</sup>lt;sup>c</sup>The rAvPAL-PEG dose may be reduced or interrupted if necessary per investigator determination.

<sup>&</sup>lt;sup>d</sup> If a subject has an NCI-CTCAE grade ≥3 hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor, the subject may be permanently discontinued from study drug.

<sup>°</sup>If the investigator determines that the NCI-CTCAE grade ≥3 hypersensitivity AE is related to administration with rAvPAL-PEG, the subject will be asked to return to the clinic within 24 hours of event onset for evaluation, including laboratory tests (chemistry, hematology, urinalysis, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE [sampling must be performed >8 hours after event onset and before the next dose of study drug], urine albumin/creatinine ratio, urinary N-methyl histamine, CRP, C3, C4, and tryptase).



# 9.1.1.3 Response to Anaphylaxis

If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and tryptase (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then be made whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose level.

For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equipment for emergency resuscitation (including epinephrine) within easy access. The subject must be observed for 30 minutes following administration due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated.

# 9.1.2 Study Stopping Criteria

If an NCI-CTCAE grade  $\geq$  3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening or required treatment to prevent a life-threatening event:

- Cyanosis or  $SpO_2 \le 92\%$
- Hypotension with SBP < 90 mm Hg (adults)
- Neurologic alteration: loss of consciousness, collapse, incontinence

Brown's severity criteria are presented in Table 9.1.2.1.

|--|

Table 9.1.2.1: Brown's Severity Criteria

| Brown's Criteria for | |
|---|---|
| Hypersensitivity Reactions | Definition |
| Mild (1) | Generalized erythema, urticaria, periorbital edema, or angioedema |
| skin and subcutaneous tissue | |
| Moderate (2) | Dyspnea, stridor, wheeze, nausea, vomiting, dizziness (pre-syncope), |
| features suggested respiratory, | diaphoresis, chest or throat tightness, or abdominal pain |
| cardiovascular, or | |
| gastrointestinal involvement | |
| Severe (3) | Cyanosis or SpO <sub>2</sub> $\leq$ 92% at any stage, hypotension (SBP $\leq$ 90 mm Hg in |
| hypoxia or neurologic | adults), confusion, collapse, loss of consciousness, or incontinence |
| compromise | |

#### 9.1.3 Dose Modifications

# 9.1.3.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events for an individual subject. Dose increases >350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.



# 9.1.3.2 Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse event (any hypersensitivity reaction as defined in Section 9.1.1). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be adjusted.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L ), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

# 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

# 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.



- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the sponsor's medical monitor. However, subjects who discontinued from study treatment early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.



- 8. Known hypersensitivity to rAvPAL-PEG necessitating early termination from a previous rAvPAL-PEG study or known hypersensitivity to any of its excipients.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

### 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study treatment should continue to perform the study tests and evaluations until study completion. For subjects who discontinue from the study, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study treatment include, but are not limited to, the following:

- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy).

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.

If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified



letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

# 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in their previous rAvPAL-PEG study. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.

### 9.4 Treatments

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies will be dosed with the same or higher dose that was administered upon completion of that study provided that there was no interruption in dosing. rAvPAL-PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be adjusted per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects may be eligible to self-administer study drug if he or she meets the following criteria:



- The subject has no cognitive impairments that may increase the safety risk of self-administration per the assessment of the investigator.
- The subject has been approved for self-administration of study drug by the sponsor's medical monitor.
- The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely.
- The subject has been provided with two epinephrine injectors and has been trained on when and how to administer it. The subject will be instructed to carry one epinephrine injector with them at all times.

Qualified study site personnel will train each eligible subject on all procedures for self-administration of study drug (vial and syringe and prefilled syringe drug products) under the supervision of the PI. Qualified study site personnel will also be required to observe the subject prepare and perform at least 1 injection prior to allowing the subject to self-administer a dose at home. The subject will see a study site nurse or home healthcare nurse in person every week or receive a telephone call from site staff to ensure that the subject continues to perform all self-administration procedures correctly, to assess adverse events, and to answer questions throughout the duration of the study. The study site nurse or home healthcare nurse will also perform the regularly scheduled assessments and procedures as outlined in Table 9.1.1 and Section 12; the subject must perform a clinic visit monthly at minimum. Training materials and other information specific to the study site personnel are provided in the Subject Self-Administration Training Materials. Prefilled syringes are dispensed to subjects only after the subject (or caregiver) has completed training and competency is demonstrated in the clinic. Additional regular refresher training occurs in the clinic, every 24 weeks, and more often as needed.

Subjects who are eligible for self-administration will be provided with a Subject Study Manual. Self-administration training materials will be provided in the Subject Study Manual to supplement the in-person training provided by the qualified study site personnel. The Subject Study Manual will include step-by-step instruction on the following:

- How to prepare and perform the injections of study drug safely.
- How to receive, track, store, prepare, and return both used and unused study drug.
- How to safely use and dispose of syringes, including prefilled syringes, used for injections of study drug.
- How to use a new syringe and vial or new prefilled syringe every time drug is administered.



- How to care for their injection site after an injection of study drug.
- How to identify an adverse reaction and how to report this reaction to the study site.
- How and when to use epinephrine injectors.
- Who to contact at the study site in case of an emergency.

The PI or the sponsor's medical monitor may request that self-administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse.

Subjects who are within the target Phe range may also be permitted to convert from weight-based dosing to fixed dosing (refer to Section 9.4.4).

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site or subject with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplying the study drug to subjects who qualify for self-administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites.

Information regarding supplying study drug to subjects who qualify for self-administration is provided in the Subject Self-Administration Training Materials.

# 9.4.2 Identity of Investigational Product (IP)

### 9.4.2.1 Product Characteristics and Labeling

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self-administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5±0.2 mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

Or

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8±0.3 mL to deliver 20 mg of rAvPAL-PEG per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8±0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

|----------|------------|---------|

Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Table 9.4.2.1.1: Prefilled Syringe Volume, Concentration, and Dose

| <b>Prefilled Syringe</b> | Volume | Concentration | Dose |
|--------------------------|--------|---------------|--------|
| Sku #1 | 0.5 mL | 5 mg/mL | 2.5 mg |
| Sku #2 | 0.5 mL | 20 mg/mL | 10 mg |
| Sku #3 | 1.0 mL | 20 mg/mL | 20 mg |

Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be eligible to transition from vial and syringe to prefilled syringe dosing. Additionally, regular refresher training on use of prefilled syringe will be provided in study clinic every 24 weeks, and more often as needed.

Subjects should convert their vial and syringe dose to prefilled syringe dose using the following table:

Table 9.4.2.1.2: Conversion from Vial and Syringe Dose to Prefilled Syringe Dose

| Daily Dose (mg)<br>Range | Daily Dose (mg)<br>Round To <sup>a</sup> | # of 2.5mg<br>Prefilled Syringe<br>Needed | # of 10mg Prefilled<br>Syringe Needed | # of 20mg Prefilled<br>Syringe Needed |
|---|---|---|---|---|
| 0 - 3.7 | 2.5 | 1 | 0 | 0 |
| 3.8 - 6.2 | 5 | 2 | | |
| 6.3 - 8.7 | 7.5 | 3 | | |
| 8.8 – 11.2 | 10 | | 1 | |
| 11.3 – 13.7 | 12.5 | 1 | 1 | |
| 13.8 – 16.2 | 15 | 2 | 1 | |
| 16.3 – 18.7 | 17.5 | 3 | 1 | |
| 18.8 – 21.2 | 20 | | | 1 |
| 21.3 – 23.7 | 22.5 | 1 | | 1 |
| 23.8 – 26.2 | 25 | 2 | | 1 |
| 26.3 – 28.7 | 27.5 | 3 | | 1 |
| 28.8 – 31.2 | 30 | | 1 | 1 |
| 31.3 – 33.7 | 32.5 | 1 | 1 | 1 |



PAL-003 A6


| Daily Dose (mg)<br>Range | Daily Dose (mg)<br>Round To <sup>a</sup> | # of 2.5mg<br>Prefilled Syringe<br>Needed | # of 10mg Prefilled<br>Syringe Needed | # of 20mg Prefilled<br>Syringe Needed |
|---|---|---|---|---|
| 33.8 - 36.2 | 35 | 2 | 1 | 1 |
| 36.3 – 38.7 | 37.5 | 3 | 1 | 1 |
| 38.8 – 41.2 | 40 | | | 2 |
| 41.3 – 44.9 | 42.5 | 1 | | 2 |
| 45 – 54.9 | 50 | | 1 | 2 |
| 55 – 64.9 | 60 | | | 3 |
| 65 – 74.9 | 70 | | 1 | 3 |
| 75 – 84.9 | 80 | | | 4 |
| 85 – 94.9 | 90 | | 1 | 4 |
| 95 – 104.9 | 100 | | | 5 |
| 105 – 114.9 | 110 | | 1 | 5 |
| 115 – 124.9 | 120 | | | 6 |
| 125 – 134.9 | 130 | | 1 | 6 |
| 135 – 144.9 | 140 | | | 7 |
| 145 – 154.9 | 150 | | 1 | 7 |

<sup>&</sup>lt;sup>a</sup> For <45 mg/day, round to nearest 2.5 mg; for ≥45 mg/day, round to nearest 10 mg.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60 600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity AE) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

For vial and syringe, drug product packaging will be identified with the lot number and expiration date and will be provided in a box labeled with the study number.



For prefilled syringe, drug product packaging will be identified with the size (2.5 mg, 10 mg, or 20 mg), lot number, and kit identification (ID). The expiration date will be available in a separate Certificate of Compliance issued for each lot.

# 9.4.3 Storage

IP must be stored at  $5 \pm 3^{\circ}$  C  $(41 \pm 5^{\circ}$  F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

Specific instructions for storage of study drug for subjects who qualify for self-administration are provided in the Subject Self-Administration Training Materials.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg (or 375 mg for subjects receiving a fixed dose).

For subjects receiving weight-based dosing, dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information presented in Table 9.4.4.1.

Table 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen

| Weight-based dose (mg/kg) | Equivalent fixed dose (mg) | Vol for 15 mg/ml concentration (ml) (vial) <sup>a</sup> |
|---|---|---|
| 0.03 | 2.5 | 0.17 |
| 0.06 | 5 | 0.33 |
| 0.12 | 10 | 0.67 |
| 0.25 | 20 | 1.33 |
| 0.5 | 40 | 2.67 |
| 1.0 | 75 | 5 |
| 2.0 | 150 | 10 |
| 3.0 | 225 | 15 |
| 4.0 | 300 | 20 |
| 5.0 | 375 | 25 |

<sup>&</sup>lt;sup>a</sup> Applies to both 1.0 and 1.3 ml withdrawal.

It is preferable that the injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff, other qualified and trained study personnel, or qualified subjects.

Information for dosing of subjects who enroll into this study after completing previous rAvPAL studies is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10.

Instructions for administration of study drug for subjects who qualify for self-administration are provided in the Subject Self-Administration Training Materials.

### 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.



Subjects will retain the same subject number used in their previous rAvPAL-PEG study.

### 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study.

## 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered by clinic staff or other qualified and trained study personnel.

Subjects may self-administer study drug at home if approved by the sponsor's medical monitor and if adequate training is provided (refer to Section 9.4).

# 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the sponsor's medical monitor must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in a previous rAvPAL-PEG study) or investigational medical device within 30 days before Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior hypersensitivity AE to rAvPAL-PEG or a PEG-containing product will be encouraged to be premedicate as outlined in Section 9.1.1. If the hypersensitivity AE worsens with a repeat injection (as determined by the Investigator in consultation with the sponsor's medical monitor) even with premedication prior to study drug


dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior hypersensitivity AE to rAvPAL-PEG or a PEG-containing product may participate in this study (refer to Section 9.3.2).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

# 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

## 9.4.10 Dose Interruption and Missed Doses

Information for dosing of subjects who enroll into this study after completing previous rAvPAL-PEG studies is provided in Section 9.1.

During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator. After a dosing interruption of ≥ four consecutive doses, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first week of dosing of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30 minutes following administration due to restarting dosing. Premedication with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to study drug should be administered following any dose interruption of ≥ four consecutive doses. NSAIDs should be given with food and may be omitted if not tolerated. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects should continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 9.1.1) during any dosing interruption.

Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study treatment per discretion of the Sponsor or Investigator (refer to Section 9.3.3).

## 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), IP returned, and IP lost or accidentally or deliberately destroyed. The PI or



designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

## 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

Subjects who qualify for self-administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials).

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

## 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator.

A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next monthly study visit. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4.

## 9.7 Efficacy and Safety Variables

#### 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1. 

|----------|------------|---------|

**Table 9.7.1.1: Summary of Laboratory Assessments** 

| Laboratory Assessment | Party Responsible for<br>Performing Test | Section in Protocol for Details |
|---|---|---|
| Clinical laboratory tests | Central laboratory | 9.7.6 |
| Antibody testing | BioMarin <sup>a</sup> or CRO | 9.7.5.2 |
| PK variables | BioMarin | 9.7.3 |
| Blood Phe concentrations | Central laboratory | 9.7.2.1 |
| Pregnancy test (urine) and sedimentation rate | Local laboratory | 9.7.6, 9.7.5.1 |
| Urinalysis | Central laboratory | 9.7.6 |

Phe, phenylalanine; PK, pharmacokinetic.

## 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, including allergy history, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

## 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

# 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. Weight will be measured at Screening and then monthly.

#### 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the Final Follow-Up (F/U) Visit or Early Termination Visit (ETV). If clinically significant

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL IgE and anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

# **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Screening, Week 48, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

# 9.7.2 Efficacy Variable

## 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn monthly, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1).

Blood Phe may be collected more often than monthly at the discretion of the Investigator should more frequent monitoring of blood Phe levels be clinically required.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Subjects enrolled in the Substudy will have additional PK sampling performed. For subjects participating in the Substudy, PK sampling will be performed as follows:

- For subjects who are administered rAvPAL-PEG once per week, plasma PK sampling will be performed pre-dose and every 24 hours thereafter (24, 48, 72, and 96 hours if possible), and then pre-dose of the next weekly dose.
- For subjects who are administered rAvPAL-PEG two or three times per week, plasma PK sampling will be performed pre-dose and every 24 hours during the longest period between doses, when possible, and then pre-dose of the next dose.
- For subjects who are administered rAvPAL-PEG four to seven times per week, plasma PK sampling will be performed pre-dose and every 12 hours during the longest period between doses, when possible, and then pre-dose of the next dose.

See Table 9.1.2 for additional details.

BioMarin will perform the analysis.

# 9.7.4 Exploratory Efficacy Variable

Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits on a monthly basis. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods



consumed for 3 consecutive days each month. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator.

# 9.7.5 Safety Variables

# 9.7.5.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 9.1.1). Female subjects with a positive serum pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.4 for details on the reporting procedures to follow in the event of pregnancy.

# 9.7.5.2 Antibody Testing

Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1). Immunogenicity assays will be performed at the time points indicated in the Schedule of Events (Table 9.1.1).

BioMarin or CRO will perform all anti-body testing, except for IgE antibodies, which will be assessed by a Contract Research Organization.

## 9.7.6 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.

All abnormal clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the abnormal result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.



PAL-003 A6


# **Table 9.7.6.1: Clinical Laboratory Tests**

| Blood Chemistry | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if applicable <sup>a</sup> |
| Alkaline Phosphatase | Hematocrit | Color | |
| ALT (SGPT) | WBC count | pH | Phenylalanine |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Sedimentation rate <sup>a</sup> |
| BUN | Differential cell count | Protein | - |
| Creatinine | | Glucose | - |
| GGT | | Spot urine albumin/creatinine ratio | Additional Unscheduled<br>Hypersensitivity Reaction<br>Visit Tests <sup>b</sup> |
| Total protein | | Nitrite | CH50 |
| Calcium | | Urobilinogen | $C_1, C_3, C_4$ |
| Sodium | | Hemoglobin | Serum tryptase level <sup>b</sup> |
| Potassium | | Bilirubin | CRP |
| Glucose | | | Urine N-methyl histamine |
| | | | Urine albumin/creatinine ratio |
| Uric acid | | | Complement Testing <sup>c</sup> |
| CO <sub>2</sub> | | | $C_3$ |
| Chloride | | | $C_4$ |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; C, complement; CH50, total hemolytic complement; CO2, carbon dioxide; CRP, C-reactive protein; GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.

<sup>&</sup>lt;sup>a</sup> To be performed by central laboratory. If urine pregnancy test is positive or equivocal, serum sample will be taken and assessed by a central laboratory.

<sup>&</sup>lt;sup>b</sup> Perform within 24 hours of event onset.

 $<sup>^{</sup>c}$  Complement  $C_3$  and  $C_4$  to be drawn at the Screening Visit and then quarterly or as needed to resolve abnormal test results.



#### 10 REPORTING ADVERSE EVENTS

#### **10.1** Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a subject administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment run-in).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The study AE reporting period is as follows: After informed consent but prior to initiation of study treatment, only SAEs associated with any protocol-imposed interventions will be reported. After informed consent is obtained and the first administration of study drug, all non-serious AEs and SAEs reporting period begins and continues until 4 weeks following the last administration of study drug or the early termination visit, whichever is longer (refer to Section 12). The criteria for determining, and the reporting of SAEs is provided in Section 10.2.

For this study, a medical device is defined as the prefilled syringe and all of the component parts. The reporting period for device-related events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe. Events assessed by the investigator as related to the device, including malfunction, injury, or medication error, will be captured into an electronic data capture system. All serious events related to the device will be reported to BioMarin Pharmacovigilance (BPV) within 24 hours using the device-related event report form and entered onto the appropriate eCRF page(s) as required.



The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or study participation is not the cause of the AE. Outcome of AEs (and resolution dates) should be documented on the appropriate CRF page(s) and in the subject's medical record unless the subject is lost to follow-up or it has been determined that the study treatment or study participation is not the cause of the AE.

The Investigator responsible for the care of the subject or qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to seriousness, which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the severity of each AE using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.

| Grade | Description |
|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life-threatening: hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL) <sup>b</sup> |
| 4 | Life threatening or debilitating: consequences; urgent intervention indicated |
| 5 | Death related to AE |

Grade 4 and 5 AEs should always be reported as SAEs.

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

<sup>&</sup>lt;sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.

|-----------------------------|
|-----------------------------|

The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly Related | The administration of the IP and the occurrence of the AE are reasonably related in time AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably Related | The administration of IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE is more likely explained by exposure to the IP than by other factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).

## **10.2** Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Is fatal.
- Is life threatening.
  - Note: Life-threatening refers to an event that places the subject at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires or prolongs inpatient hospitalization.
- Results in persistent or significant disability or incapacity.
- Is a congenital anomaly or birth defect in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Important medical events or reactions that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes above should also usually be considered serious.



For this protocol, anaphylaxis per NIAID/FAAN criteria for the clinical diagnosis of anaphylaxis is designated as an AE of special interest (serious or nonserious and irrespective of severity) to facilitate rapid reporting and sponsor review. All occurrences of anaphylaxis per NIAID/FAAN criteria will be reported to the sponsor within 24 hours of the site becoming aware of the event using the SAE form. Severity and serious criteria (if applicable) should be reported on the SAE form.

The reporting period for SAEs related to protocol imposed interventions begins after informed consent is obtained, the reporting period for all SAEs begins after first dose of study drug and continues until 4 weeks following the last administration of study drug or End of Treatment Visit. The reporting period for Serious Device Related Events begins after first dose of study drug and ends with the last administered dose.

All SAEs (including serious device-related events), whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form or device Report Form to BioMarin Pharmacovigilance (BPV). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the subject's medical record.

For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).

At the last scheduled visit, the Investigator should instruct each subject to report any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study treatment.

The Investigator should notify the study Sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior study treatment. The Sponsor should also be notified if the Investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that participated in this study.



Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

## 10.3 Pregnancy

Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. The reporting period for pregnancies begins with informed consent and continues until 4 weeks following the last study drug dose. In addition, pregnancy in a subject is also reported on the End of Study CRF. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution to BPV in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

## 10.4 Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "...in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours.

Examples of situations that may require urgent safety measures include discovery of the following:

• Immediate need to revise the IP administration (i.e., modified dose amount or frequency not defined in protocol).



- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.

# 10.5 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the Sponsor's Medical Office sponsor's medical monitor r any AEs for which the issue of seriousness is unclear or questioned. Contact information for the sponsor's medical monitor is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:

Fax:

E-mail:



#### 11 APPROPRIATENESS OF MEASUREMENTS

# 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

# 11.2 Diet Diary

A 3-day diet diary will be issued to subjects for completion and will be brought to clinic on a monthly basis for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6.



#### 12 STUDY PROCEDURES

## 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

# 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Chest X-ray
- 12-lead ECG
- Clinical laboratory tests (including spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis)
- Complement C<sub>3</sub> and C<sub>4</sub>
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in a previous rAvPAL-PEG study, these assessments may be the same as those used for the last visit of the previous study, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done predose unless



otherwise specified. Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done daily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

# 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator)

## 12.3.2 Weekly Telephone Visit

Subjects should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit:

- Injection-site self inspection (previous and current injection site)
- Assessment of AEs
- Concomitant medications



• Confirmation of dose level, frequency, and study drug administration

#### 12.3.3 Substudy Visits

For subjects participating in the PK substudy, refer to Section 9.7.3 and Table 9.1.2.

#### 12.3.4 Monthly Visits (Week 4, 8, 12, etc)

Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Beginning with Week 4, monthly visits must be performed in the clinic. The following study activities will be performed:

- Vital signs
- Weight
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) For safety reasons, this test must be performed prior to the chest X-ray.
- Chest x-ray (Week 48 visit only)
- Assessment of AEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.)
- Prefilled syringe self-administration training (to be performed prior to subjects transitioning from vial and syringe drug product to prefilled syringe drug product).
- If additional training is needed on days subsequent to the monthly visit, additional clinic visit(s) or HHRN may be used.

## 12.3.5 Quarterly Visits (Week 12, 24, 36, etc)

Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Beginning with Week 12, quarterly visits consist of all monthly (Section 12.3.4) activities listed above as well as the additional study activities listed below:



- Physical examination
- Complement C<sub>3</sub> and C<sub>4</sub>
- Sedimentation rate
- PK sample
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Prefilled syringe refresher training (every 24 weeks only)

# 12.3.6 Unscheduled Hypersensitivity Reaction Visit

Subjects who have an NCI-CTCAE grade  $\geq$  3 hypersensitivity reaction after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 24 hours) the reaction.

- Vital signs
- Clinical laboratory tests
- Urine/albumin creatinine ratio
- CRP, CH50, C1, C3, and C4
- Urine N-methyl histamine
- Serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only (performed > 8 hours after event onset)
- Serum tryptase level
- Skin biopsy (optional; affected and not affected area; to be performed within 1 week of the reaction)
- Assessment of AEs
- Concomitant medications

Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects may resume study drug administration per the discretion of the Principal Investigator and the sponsor's medical monitor.

#### 12.4 Early Termination Visit

The Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug. Subjects who terminate from study treatment early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion.



Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)

### 12.5 Final Follow-up Visit

The final follow-up (F/U) Visit will occur 4 weeks after the final dose of study drug.

The following study activities will be performed at the F/U Visit:

- Physical examination
- Vital signs, including weight
- 12-lead ECG
- Clinical laboratory tests



- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Final Follow-up Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)



## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

## 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF).

The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics of vital signs, physical examination results, ECG results, and X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

## 14.3 Pharmacokinetic Analysis

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F). Should 



data become available from previous rAvPAL-PEG studies that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

# 14.3.1 Pharmacokinetic Substudy Analysis

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored. This substudy has been completed as of 20 December 2013.

## 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the SAP) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis.

Details regarding exploratory analyses will be provided in the Statistical Analysis Plan.

## 14.5 Determination of Sample Size

Subjects who participated in previous rAvPAL-PEG studies may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

## 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.



#### 14.7 Interim Analyses

Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

## 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.



# 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Assess the effect and relevance of new external evidence.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.2.
- Make recommendations to the BioMarin concerning continuation or termination of the study or other study modifications based on observations.



## 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment, unless the executed Clinical Trial Agreement between BioMarin and the institution of the investigator specifies otherwise. If the subject has followed the Investigator's instructions, BioMarin may pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.



#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.



#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (e.g., subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.



## 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages their publication in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Study Agreement between BioMarin and the PI.



#### 21 REFERENCES

Armstrong, JK, Hempel, G, Koling, S, Chan, LS et. al. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007

Brown, SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 114[2], 371-376. 2004

Chen, AM, Scott, MD. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001

Davis, S, Abuchowski, A, Park, YK, Davis, FF. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981

Fisch, RO. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000

Gamez, A, Wang, L, Sarkissian, CN, Wendt, D et. al. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007

Ganson, NJ, Kelly, SJ, Scarlett, E, Sundy, JS et. al. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006

Guttler, F, Azen, C, Guldberg, P, Romstad, A et. al. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003

Harris, JM, Chess, RB. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003

Huttenlocher, PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000

Judge, A, McClintock, K, Phelps, JR, Maclachlan, I. Hypersensitivity and loss of disease site targeting caused by antibody responses to PEGylated liposomes. Mol Ther 13[2], 328-337. 2006

Kaufman, S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989

Koch, R, Hanley, W, Levy, H, Matalon, K et. al. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003



Lapis. Long-term Correction of PKU in the Pahenu2 Mouse by Mutant and Chemically Modified Forms of Phenylalanine Ammonium Lyase. ASHG 57th Annual Meeting The American Society of Human Genetics) 2007.

Lee, PJ, Lilburn, M, Baudin, J. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003

Levy, HL. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003

Matalon, R, Surendran, S, Matalon, KM, Tyring, S et. al. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003

Richter, AW, Akerblom, E. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983

Richter, AW, Akerblom, E. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984

Rouse, B, Azen, C. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004

Sampson, HA, Munoz-Furlong, A, Campbell, RL, Adkinson, NF, Jr. et. al. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol 117[2], 391-397. 2006

Scott, MD, Murad, KL, Koumpouras, F, Talbot, M et. al. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997

Scriver, CR, Kaufman. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-1724.

Walter, JH, White, FJ, Hall, SK, MacDonald, A et. al. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002

Webster, R, Didier, E, Harris, P, Siegel, N et. al. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007



# 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.

Date



#### 23 SIGNATURE PAGE

Investigator

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003, Amendment 6

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

Signature

| Printed name: | |
|---------------------------|-----------|
| Accepted for the Sponsor: | |
| | 30 Oct 20 |



PAL-003 A6


# 24 PROTOCOL AMENDMENT MAJOR TEXT REVISIONS

| Section no./Title | Text Revisions |
|---|---|
| | Rationale #1: Eligibility for receiving open-label drug in current or extension study |
| 9.1 Overall Study Design<br>and Plan | Subjects who participate in this study will be required to transition into a Phase 3 study (165-302) if weekly doses of rAvPAL PEG are between 70 mg/week and 350 mg/week (inclusive) provided that doses of rAvPAL PEG have been stable (ie, no major change in dose for at least 4 weeks). Subjects who meet these criteria must be transitioned from PAL 003 to Study 165-302 provided they meet the 165-302 study eligibility criteria. Subjects who are eligible for Study 165-302 but do not transition into 165-302 will be withdrawn from this study. The PAL 003 study will continue until BMN 165 is approved by the FDA for marketing in the United States or until the sponsor terminates further development of this drug for treatment of PKU. |
| | Rationale #2a-c: Revisions to Stopping Criteria, AEs of special interest |
| 9.1.1.1 Individual Stopping<br>Criteria | 9.1.1.1 Individual Stopping Criteria Subjects who have an NCI CTCAE grade ≥ 3 hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug. |
| 9.1.1.2 Dosing in Response<br>to Hypersensitivity Adverse<br>Events | 9.1.1.2 Dosing in Response to Hypersensitivity Adverse Events Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG. Dosing instructions are presented in Table 9.1.1.2.1 and are regardless of previous occurrence: PLEASE SEE TABLE 9.1.1.2.1 AT THE END OF SECTION 24 |
| | 9.1.2 Study Stopping Criteria If an NCI-CTCAE grade ≥ 3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening |

|----------|------------|---------|
|----------|------------|---------|

| | or required treatment to prevent a life-threatening event: |
|---|---|
| | • Cyanosis or $SpO_2 \le 92\%$ |
| | • Hypotension with SBP < 90 mm Hg (adults) |
| | Neurologic alteration: loss of consciousness, collapse, incontinence |
| | Brown's severity criteria are presented in Table 9.1.2.1. |
| | PLEASE SEE TABLE 9.1.2.1 AT THE END OF SECTION 24 |
| 9.1.3 Safety Assessment | 9.1.3 Safety Assessment Criteria |
| Criteria | If an individual subject exhibits toxicity of a treatment emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, that subject will have dosing halted until the toxicity resolves. The subject's data will be evaluated by the Principal Investigator (PI) and the Sponsor's Medical Officer, and a decision will then be made whether to discontinue the subject from the study treatment, restart dosing at the same dose level, or restart dosing at a lower dose level. |
| 9.1.4 Stopping Criteria | 9.1.4 Stopping Criteria |
| | If 2 or more subjects at a dose level exhibit toxicity of a treatment emergent CTCAE grade 3 or greater or a systemic reaction that is assessed as related to treatment with study drug, further dosing of subjects at that dose level will evaluated and a safety assessment will be completed. In addition, the Food and Drug Administration (FDA) may be notified of this occurrence if appropriate. |
| 10.2 Serious Adverse | For this protocol, anaphylaxis per NIAID/FAAN criteria for the clinical diagnosis of anaphylaxis is designated as an AE of special interest |
| Events | (serious or nonserious and irrespective of severity) to facilitate rapid reporting and sponsor review. All occurrences of anaphylaxis per NIAID/FAAN criteria will be reported to the sponsor within 24 hours of the site becoming aware of the event using the SAE form. Severity and serious criteria (if applicable) should be reported on the SAE form. |
| | Rationale #3: |
| | Resumption of drug after anaphylaxis |
| 9.1.1.3 Response to<br>Anaphylaxis | 9.1.1.3 Response to Anaphylaxis If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and |

|---|---|---|
| anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose le For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equip emergency resuscitation (including epinephrine) within easy access. The subject must be observed for 30 minutes followin due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and NSAIDs 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption should be given with food and may be omitted if not tolerated. | | monitor, and a decision will then be made or restart dosing at a lower dose level. stered in a clinic setting with equipment for observed for 30 minutes following administration onist, H2 antagonist, and NSAIDs approximately |
| | Rationale # 4a, 4b: Safety precautions added regarding premedication and epinephrine injectors | |
| 7.4.3 Management of Hypersensitivity Reactions | Because of the small potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection. Subject should be pre-medicated with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated. Subjects who qualify for self-administration of study drug will be provided with emergency resuscitation are trained to recognize a serious hypersensitivity AEs and how to respond. Additionally, subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (Section 9.4). Refer to Section 9.1.1.3 for instructions (refer to Section 9.4 and the Subject Self Administration Training Materials)-regarding resumption of study drug following resolution of symptoms consistent with a clinical diagnosis of anaphylaxis per National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria (Sampson, H. A., et al, 2006, J Allergy Clin Immunol). • Administration of additional symptomatic treatment (eg, acetaminiophen or ibuprofen). An allergy and/or immunology consultation should be sought if necessary. Information regarding the management of local skin, large local skin, and systemic reactions is provided in Section 9.11. Detailed instructions | |
| 9.1.1 Response to Hypersensitivity Adverse Events | Subjects who quali | nt of Local and Systemic Reactions to rAvPAL PEG fy for self administration of study drug will be provided with informati reactions (refer to the Subject Self Administration Training Materials). |
| | 9.1.1 Response to Hypersensitivity Adverse Events Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) | |



and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. NSAIDs should be given with food and may be omitted if not tolerated.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality (Section 9.1.1.3). Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

# 9.1.1.1 Subjects Who Have Had Previous Hypersensitivity Reactions to rAvPAL PEG or a PEG containing Product

Subjects who had a previous systemic reaction to rAvPAL PEG or a PEG containing product that warranted early termination from a previous rAvPAL PEG study are excluded from participation in this study. Subjects who have had a previous local skin reaction to rAvPAL PEG in a previous rAvPAL PEG study are eligible to participate in this study. Subjects who have had a previous reaction and are deemed eligible for participation must be premedicated orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing for the remainder of the study. The premedication dosage will be standard. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable). Subjects may develop systemic, large local skin, or local skin reactions after enrollment in PAL 003. Refer to Section 9.1.1.2 for definitions of systemic and local skin reactions. For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and 9.1.1.3.1.

# 9.1.1.2 Definition of Reaction and Hypersensitivity Reactions to rAvPAL PEG Administered Subcutaneously

During Study PAL 003, subjects may experience hypersensitivity reactions to rAvPAL PEG. The hypersensitivity reactions are defined as follows:

#### Local skin reaction:

• Skin signs or symptoms in 1 affected primary location, ie, hives, wheals, or swelling or an area of erythema, redness, induration, pain, or itching at or near the site of injection.

#### Large local skin reaction:

• Skin signs or symptoms, ie, hives, wheals, or swelling or an area of erythema, redness, or induration with pain or itching that extends beyond the site of injection by approximately 6 inches (15 cm) and/or signs or symptoms that are not contiguous to the injection site. These may be associated with a low risk of systemic symptoms or anaphylaxis upon re exposure and, therefore, will be managed as a systemic reaction when not contiguous to the injection site.




Systemic reaction (including generalized skin symptoms):

• Skin and non skin signs or symptoms in more than 1 affected primary location, ie, cutaneous reaction in more than 1 area and/or anaphylaxis or any other generalized symptoms, such as hypotension, angioedema or the involvement of other organ systems, eg, respiratory, cardiovascular, gastrointestinal, neurological; and/or a fever attributed to treatment with rAvPAL PEG (≥ 100.4°F or ≥ 38°C).

For management of hypersensitivity reactions that occur during this study, refer to Section 9.1.1.3 and Figure 9.1.1.3.1.

#### 9.1.1.3.1 Local Skin Reactions

All subjects who experience a local skin reaction during this study may be premedicated orally with acetaminophen and/or non sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non sedating premedications prior to coming to clinic) for all future study doses. Recommended premedications are acetaminophen and/or non-sedating antihistamine. The dosage will be standard. Subjects must be accompanied by a designated driver (if applicable) because antihistamines can cause drowsiness. Symptoms of local reactions may be treated with local application of ice and non-sedating oral and/or topical antihistamines and/or topical steroids (refer to Section 7.4.3).

If the local skin reaction worsens with a repeat injection (as determined by the Investigator in consultation with the Sponsor's Medical Officer) even with premedication prior to study drug dosing, the subject must be withdrawn from study treatment.

### 9.1.1.3.2 Large Local Skin Reactions

Large local skin reactions (refer to Section 9.1.1.2 for a definition) may or may not be contiguous to the rAvPAL PEG injection site, and subjects with either type of large local skin reaction may continue dosing if the skin symptoms have resolved and no other symptoms have developed. Subjects will be encouraged to premedicate orally with acetaminophen and/or non sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non sedating premedications prior to coming to clinic) for all future study doses.

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.3).

9.1.1.3.2.1 Large Local Skin Reactions Contiguous to Injection Site




Subjects who develop a large local skin reaction contiguous to the injection site after administration of rAvPAL PEG or to rAvPAL PEG or a PEG containing product may remain in the study if the skin symptoms have resolved and no other symptoms have developed. For the remainder of the study, subjects will be encouraged to premedicate orally with acetaminophen and/or non-sedating antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming to clinic) for all future study doses. Because antihistamines can cause drowsiness, it may be administered only if the subject is accompanied by a designated driver (if applicable).

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.3).

### 9.1.1.3.2.2 Large Local Skin Reactions Not Contiguous to Injection Site

Large local skin reactions that are not contiguous to the injection site may be associated with a low risk of systemic symptoms or anaphylaxis upon re-exposure to rAvPAL PEG and, therefore, will be managed as a systemic reaction (refer to Section 9.1.1.3.3). An example of a large local reaction that is not contiguous to the injection site is if an injection took place in the right upper arm and there are lesions beyond the elbow joint in the right forearm or lesions beyond the shoulder joint on the right trunk.

Symptoms of large local skin reactions may be treated with local application of ice and topical, oral, or IV antihistamines and/or steroids as needed (refer to Section 7.4.3).

### 9.1.1.3.3 Systemic Reactions

Subjects who experience a systemic reaction (refer to Section 9.1.1.2 for a definition) after administration of rAvPAL PEG must stop further administrations of rAvPAL PEG and must immediately return to the clinic for safety assessments. Subjects who experience generalized skin symptoms are included in this category. Immediately after the systemic reaction (within 24 hours), subjects with generalized skin symptoms must have additional assessments performed for safety (ie, Unscheduled Hypersensitivity Reaction Visit): serum antibodies (anti PAL IgG, anti PAL IgM, anti PEG IgG, anti PEG IgM, anti rAvPAL PEG IgE, anti rAvPAL PEG neutralizing antibodies); serum tryptase level (it is recommended that this sample be drawn immediately after reaction); urine albumin/creatinine ratio; urine N methyl histamine; CRP, CH50, C<sub>1</sub>, C<sub>3</sub>, and C<sub>4</sub>; skin biopsy (optional; affected and not affected area; to be performed within 1 week of reaction); and clinical laboratory tests (urinalysis, chemistry, hematology; refer to Figure 9.1.1.3.1.

Following the reaction, subjects will be required to complete the assessments of the Unscheduled Hypersensitivity Reaction visit, including assessment of IgE. If a subject presents with a clinical diagnosis of anaphylaxis, further dosing will be held while laboratory evaluation of IgE, as part of the Unscheduled Systemic Reaction Visit, is performed. Subjects may resume study drug administration per the discretion of the Principal Investigator and the Sponsor's Medical Officer; however, if subject was dosing at home, they will be required to come into

| BIO | $\vee$ | A | R | N | 8 |
|-----|--------|---|---|---|---|
|-----|--------|---|---|---|---|


| | the clinic for at least 1 week. |
|---|---|
| | rAvPAL PEG administration will resume at the next lowest dose level. Restarting of rAvPAL PEG administration following a systemic |
| | reaction must be performed in the clinic for the first week of resumed dosing. Subjects will be encouraged to premedicate orally with |
| | acetaminophen and/or antihistamines 1-2 hours prior to study drug dosing (subjects may take non-sedating premedications prior to coming |
| | to clinic) for all future study doses. Additionally, subjects must be closely monitored for 30 minutes following every administration of |
| | study drug. Because antihistamines may cause drowsiness, the subject must be accompanied by a designated driver (if applicable). |
| | If blood Phe concentrations are not 60 600 µmol/L following 1 week of daily administration at the lowered dose cohort and there is no |
| | further evidence of toxicity (ie, another systemic reaction attributed to rAvPAL PEG administration or clinically significant abnormal |
| | laboratory test results), the subject may be administered the next highest dose level in the clinic per the allowable dose increases outlined in |
| | Section 8.1.2. Subjects will be encouraged to premedicate orally with acetaminophen and/or antihistamines 1 2 hours prior to study drug |
| | dosing (subjects may take non sedating premedications prior to coming to clinic) for all future study doses. Additionally, subjects must be |
| | closely monitored for 30 minutes following every study drug administration. Because antihistamines may cause drowsiness, the subject |
| | must be accompanied by a designated driver (if applicable). |
| 9.4.10 Dose Interruption | During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator. |
| and Missed Doses | Subjects who miss more than 2 consecutive weekly doses (weekly dosing schedule) or 3 consecutive daily doses (daily dosing schedule) |
| | for whatever reason may continue participation in this study. After a dosing interruption After a dosing interruption of ≥ four consecutive |
| | doses, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the |
| | dosing interruption. The first dose of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject |
| | must be observed for 30 minutes following administration due to restarting dosing. Premedication with H1 antagonist, H2 antagonist, and |
| | non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to study drug should be administered following any |
| | dose interruption of ≥ four consecutive doses. NSAIDs should be given with food and may be omitted if not tolerated. A follow-up |
| | telephone call |
| 9.1 Overall Study Design | Subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (refer to |
| and Plan | <u>Section 9.4).</u> |
| 9.4 Treatments | The subject has been provided with two epinephrine injectors and has been trained on when and how to administer it. The subject will be |
| | instructed to carry one epinephrine injector with them at all times. |
| | Rationale #5: |
| | Information tracking system for device malfunction |

| 10111 | |
|---|---|
| 10.1 Adverse Events | For this study, a medical device is defined as the prefilled syringe and all of the component parts. The reporting period for device-related |
| | events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe. |
| | Events assessed by the investigator as related to the device, including malfunction, injury, or medication error, will be captured into an |
| | electronic data capture system. All serious events related to the device will be reported to BioMarin Pharmacovigilance (BPV) within 24 |
| hours using the device-related event report form and entered onto the appropriate eCRF page(s) as required. | |
| | Rationale #6: |
| | Changes to antibody assessment samples at Hypersensitivity Reaction Visit |
| Table 9.1.1 footnote m | For unscheduled hypersensitivity reaction visit, draw serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only; sampling must be |
| | performed > 8 hours after event onset and before the next dose of study drug. |
| 9.1.1.3 Response to | Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if |
| Anaphylaxis | applicable) and include anti-rAvPAL IgE and anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before |
| | the next dose of study drug) |
| 12.3.6 Unscheduled | Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-IgE and anti-rAvPAL-PEG IgE, |
| Hypersensitivity Visit | and anti-rAvPAL PEG neutralizing antibodies only (performed > 8 hours after event onset) |
| | Rationale #7: |
| | Prefilled syringe instructions and training |
| 9.1 Overall Study Design | Additional information is provided in the Subject Self-Administration Training Materials. Additional training will be provided and |
| and Plan | demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed. |
| Table 9.1.1 footnote q | Initial training on the use of prefilled syringe occurs at the next monthly visit and each subsequent day after transition until (in clinic or by |
| Table 9.1.1 footnote q | Initial training on the use of prefilled syringe occurs at the next monthly visit and each subsequent day after transition until (in clinic or by HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer |
| Table 9.1.1 footnote q | |
| Table 9.1.1 footnote q 9.4 Treatments | HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer |
| • | HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter. |
| • | HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter. Prefilled syringes are dispensed to subjects only after the subject (or caregiver) has completed training and competency is demonstrated in |
| 9.4 Treatments | HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter. Prefilled syringes are dispensed to subjects only after the subject (or caregiver) has completed training and competency is demonstrated in the clinic. Additional regular refresher training occurs in the clinic, every 24 weeks, and more often as needed. |
| 9.4 Treatments 9.4.2.1 Product | HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter. Prefilled syringes are dispensed to subjects only after the subject (or caregiver) has completed training and competency is demonstrated in the clinic. Additional regular refresher training occurs in the clinic, every 24 weeks, and more often as needed. Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be |

|------------------------------|--|
|------------------------------|--|

| | Revision to length of observed dosing after dose interruption |
|---|---|
| 12.5 Final Follow-up Visit | Rationale #10: |
| Table 9.1.1 Schedule of Events | Final F/U Visit: 1 week 4 weeks after final dose |
| | Rationale #9:<br>Change to follow-up visit schedule |
| Section 9.1 Overall Study<br>Design and Plan | The subject has completed the study through the Month 86 98 visit. |
| | Rationale #8: Study duration extended |
| 12.3.4 Monthly Visits | <ul> <li>Prefilled syringe self-administration training (to be performed prior to subjects transitioning from vial and syringe drug product to prefilled syringe drug product).</li> <li>If additional training is needed on days subsequent to the monthly visit, additional clinic visit(s) or HHRN may be used.</li> </ul> |
| Characteristics and Labeling | increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60 600 µmol/L), as well as any adverse events (any hypersensitivity AE) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60 -600 µmol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses. For vial and syringe, drug product packaging will be identified with the lot number and expiration date and will be provided in a box labeled with the study number. For prefilled syringe, drug product packaging will be identified with the size (2.5 mg, 10 mg, or 20 mg), lot number, and kit identification (ID). The expiration date will be available in a separate Certificate of Compliance issued for each lot. |
| 9.4.2.1 Product | Drug rAvPAL PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be |
| | PLEASE SEE THE DOSE CONVERSION TABLE AT THE END OF SECTION 24 |
| | Subjects should convert their vial and syringe dose to prefilled syringe dose using the following table: |

|----------|------------|----------|

| Section 9.1 Overall Study<br>Design and Plan | The first dose week of dosing will be administered in the clinic |
|---|---|
| Section 9.4.10 Dose<br>Interruption and Missed<br>Doses | The first dose week of dosing of rAvPAL- PEG following a dose interruption should be administered in a clinic setting |
| | Rationale #11: |
| | Inspection of injection site procedure deleted |
| Table 9.1.1 Schedule of | Table: Injection site inspection |
| Events and footnote | Footnote: Subjects must have AEs and concomitant medications assessed and an injection site inspection performed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. |
| 12.3 Treatment period | Subjects must have AEs and concomitant medications assessed and an injection site inspection performed whenever dose is administered |
| 12.3.4 Monthly visits (Week 4, 8, 12, etc) | even if the administration does not coincide with a scheduled clinic visit. |
| 12.3.5 Quarterly Visits (Week 12, 24, 36, etc) | |
| 12.3.4 Monthly visits<br>(Week 4, 8, 12, etc) | Injection site inspection (previous and current injection site) |
| 12.3.1 Day 1 (Week 1) | Injection site inspection (postdose) |
| 12.3.6 Unscheduled<br>Hypersensitivity Reaction<br>Visit | Injection site inspection |
| 12.4 Early Termination Visit 12.5 Final Follow-up Visit | Injection site inspection (previous injection site) |
| Table 9.1.1 Schedule of | Table: Injection site inspection |

| BIOMARIN <sup>®</sup> PAL-003 A6 | Page 104 |
|----------------------------------|----------|
|----------------------------------|----------|

| Events and footnote | Footnote: Subjects must have AEs and concomitant medications assessed and an injection site inspection performed whenever dose is |
|---|---|
| | administered even if the administration does not coincide with a scheduled clinic visit. |
| | Rationale #12: |
| | The criteria for subject eligibility to self-administer study drug has been revised |
| 9.4 Treatments | <ul> <li>The subject is on a stable dosing regimen for 2 weeks (ie, the subject has demonstrated a blood Phe level within 60-600 μmol/L).</li> </ul> |
| | <ul> <li>The subject has not experienced any CTCAE Grade 3 or higher adverse event.</li> </ul> |
| | The subject has not experienced any hypersensitivity reaction to rAvPAL PEG for at least 4 weeks. |
| | Rationale #13: |
| | Revision and update to the rAvPAL-PEG immunogenicity profile; additional information characterizing specific antibody |
| | responses detected in subjects |
| 7.4.2 Immunologic | 7.4.2 Toxicity Due to an Immunologic Reaction Response |
| Response | The active drug substance in rAvPAL-PEG is a bacterial protein, and as such, it is expected that it may elicitelicits immune recognition and |
| | subsequent antibody responses. Epitopes that play a role in Antibody epitopes on the immune response may protein are expected to be rendered at |
| | least partially inaccessible by PEGthe extensive PEGylation on the drug (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have |
| | shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, |
| | BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model, although PEGylationbut does not |
| | eliminate antibody formation. Although PEGylation of rAvPAL may have a significant effect on reducing likely reduces the |
| | immunogenicity antigenicity of the molecule, it is reasonable to expect that some 100% of individuals may exhibit exposed to rAvPAL-PEG develop antibodies against rAvPAL. |
| | <u>Drug-specific</u> immune responses <del>upon exposure</del> can range from clinical irrelevance to the causing serious hypersensitivity AEs (such as |
| | anaphylaxis) and may reduce efficacy due to antibody-mediated drug. These immune responses may be clinically irrelevant, cause symptoms of |
| | various degrees, clearance or lead to antibody neutralization of biological enzymatic activity. Subjects participating in clinical trials will be |
| | monitored closely with specific antibody titers sedimentation rates, and complete blood counts (CBCs). |
| | As of May 2012, a total of 70 subjects have been administered rAvPAL PEG in the single dose, Phase 1 study (PAL 001) and in the repeat |
| | dosing Phase 2 studies (PAL 002, PAL 004, and PAL 003). The dose levels in the repeat dosing studies range from 0.001 to 5.0 mg/kg/week |
| | administered in various frequencies (including 5 days a week). The most clinically significant AEs have been hypersensitivity reactions that have |
| | led to dosing interruptions and reductions. Most of the hypersensitivity reactions have been nonserious and mild to moderate in severity. |

A total of 4 SAEs have been reported in the previous rAvPAL PEG studies. Of these 4 SAEs, 3 have been reported as related to rAvPAL PEG. Two of the study drug related SAEs occurred in Study PAL 001. Both of these SAEs occurred in subjects in the lower dose cohorts: an SAE of hypersensitivity reaction in a subject in the 0.001 mg/kg cohort and an SAE of anaphylactic reaction (urticaria) in a subject in the 0.01 mg/kg cohort. Neither SAE was severe or resulted in discontinuation from the study, and both of the SAEs resolved. There were no SAEs in subjects in the higher dose cohorts (0.03 mg/kg and 0.1mg/kg) in PAL 001. The third study drug related SAE (angioedema) occurred in a subject in Study PAL 004. The fourth SAE (urticaria, dehydration) was reported as not related to study drug and occurred in a subject in Study PAL 002. There have been no reports of anaphylaxis for any subject treated with rAvPEG PAL (as of January 2012).

Subjects who have a systemic clinical reaction at any time during this study may undergo a series of assessments to monitor safety, including assessment of complements, C reactive protein (CRP), erythrocyte sedimentation rate (ESR), and IgE antibodies. Reintroduction of rAvPAL PEG dosing after a reaction will depend on clinical assessments and available laboratory data, such as chemistry and urine studies, to ensure that there has been no end organ damage prior to resuming treatment with rAvPAL PEG. As of May 2012, antibody titers, including positive IgE titers, have not been predictive of future clinical reactions when dosing with rAvPAL-PEG. Additionally, subjects may be premedicated to prevent or mitigate risk of hypersensitivity reactions (refer to Section 9.1.1.3.3).

PEG itself is considered nonimmunogenic Historically, PEG was thought to be nonimmunogenic (Davis, 1981, Clin. Exp. Immunol.), (Harris, 2003, Nat. Rev. Drug Discov.); however, repeated studies have found that subcutaneous (SC) and intravenous exposure to PEG can induce anti PEG antibodies (Harris, 2003, Nat. Rev. Drug Discov.) however, antibodies against PEG may form when PEG is bound to compounds. (Richter, 1983, Int. Arch. Allergy Appl. Immunol.). In some instances, development of such antibodies did not result in significant clinical effects in humans (Richter, 1984, Int. Arch. Allergy Appl. Immunol.). In some instances, development of such antibodies did not result in any significant clinical effects in humans. However, PEG antibody responses were associated with hypersensitivity reactions to PEGylated liposomes (Judge, 2006, Mol. Ther.). In some individuals, anti PEG antibodies may be pre-existing due to previous exposure to PEG in other products. Anti PEG antibodies have also been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res. Ther.). Administration of rAvPAL PEG may lead to anti PEG antibody formation, and the duration of this possible effect is not known. Subjects in the Phase 2 rAvPAL PEG studies have developed both anti PEG IgM and anti PEG IgG antibodies. Antibody formation may limit a subject's future ability to be treated with other PEG containing (eg, Depo Provera) or PEGylated (eg, PEG interferon) injectable drugs. It is therefore recommended that any PEG containing injectable drug administered to subjects after completion of this study be done under medical observation.

#### **Systemic Skin Reactions**

Two out of 25 subjects who were enrolled in Study PAL 001 and received the protocol defined single dose of rAvPAL PEG reported systemic skin reactions (generalized skin rash) that were attributed to treatment with study drug. One subject received a single dose of 0.001 mg/kg rAvPAL PEG, and the other subject received a single dose of 0.01 mg/kg rAvPAL PEG. One of these events was reported as serious, and the other was reported as nonserious; both events were reported following administration of Depo Provera injections (medroxyprogesterone injection), an injectable contraception. These allergic reactions are thought to be related to the PEG molecules that are found in both the study drug, rAvPAL-


PEG, and Depo Provera. These reactions are not likely to be experienced concurrent with other birth control medications.

The 2 subjects were administered study drug during PAL 001 and then experienced an allergic reaction following an injection of Depo Provera. The symptoms of the reactions were hives on the arms and legs and difficulty breathing. The symptoms for both subjects resolved within 1 day following treatment with medication, including the antihistamine Benadryl (diphenhydramine). Both subjects were examined by an allergy specialist after they completed participation in PAL 001. A skin prick test with Depo Provera was administered as part of this examination. One subject had a mild allergic reaction to the test; however, no further reactions or complications were reported following subsequent administration of a full dose of Depo Provera. Upon study completion, the subject continued to receive regular doses (every 3 months) of Depo Provera, and no further reactions were reported. The second subject also had a positive reaction to Depo Provera following administration of the skin prick test. When a subsequent full dose of Depo Provera was administered, developed hives, itching, and chills. The subject's symptoms resolved within 1 day of taking medication prescribed by an allergist. See Section 7.2.1 for the results from Study PAL 001.

The active drug substance in rAvPAL PEG is a bacterial protein that may elicit immune responses, such as urticaria, bronchospasm, itching, anaphylaxis, and others. The results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys indicated the formation of anti-rAvPAL antibody titers that did not correspond with observations of injection site reactions. Quantitation of anti-PEG titers were not assessed in the chronic repeat dose studies in the rat and monkey. Although results from nonclinical studies of rAvPAL-PEG conducted in rats and cynomolgus monkeys did not indicate signs of immune mediated toxicities, it is possible that the physio-chemical properties of rAvPAL-PEG may induce immunologic sensitization to the protein rAvPAL and to PEG in humans. It is currently unknown whether administration of PEG containing drugs, such as Depo Provera, has a sensitizing effect to PEG in rAvPAL-PEG when administered in humans. Because the exact basis for these reported events and their duration is not known, the use of PEG containing injectable drugs prior to, during, and after this study is prohibited as a precautionary measure (refer to Section 9.3.2 and Section 9.4.8).

Subjects participating in the Phase 2 clinical studies have been monitored closely for anti-drug immunogenicity (anti-rAvPAL immunoglobulin G [IgG], anti-rAvPAL IgM, anti-PEG IgM, anti-PEG IgG, neutralizing antibodies that inhibit PAL enzymatic activity, anti-rAvPAL IgE, and anti-rAvPAL-PEG IgE), complements, C-reactive protein (CRP), ESR, and complete chemistry. All subjects treated with rAvPAL-PEG in the Phase 2 clinical trials developed antibodies against the PAL protein. Anti-rAvPAL IgM antibodies were first detected within 2-3 weeks of treatment initiation and anti-rAvPAL IgG antibodies were detected within 2-3 months. The anti-rAvPAL IgG response generally peaked by 3-5 months and was sustained in all subjects. Neutralizing antibodies (NAb) capable of inhibiting enzymatic activity were detected in a minority of subjects 2-3 months after treatment initiation. The timing of the NAb response suggests these antibodies may be a component of the anti-rAvPAL IgG response. It is expected that the centralized location of the PAL active site, within the tetrameric structure, makes it difficult for antibodies to bind and inhibit enzymatic activity. In addition, anti-PAL antibody binding is likely sterically hindered by the extensive PEGylation. The majority of treated subjects also developed a transient anti-PEG antibody response. The anti-PEG response was comprised of IgM and IgG isotypes. In general, anti-PEG antibodies were no longer detected after 5-6 months of treatment. This type of transient antibody response is typical of T cell-independent type 2 (TI-2) responses.

|----------|------------|----------|
|----------|------------|----------|

The majority of immune-mediated AEs experienced in subjects treated with rAvPAL-PEG in the Phase 2 studies are believed to be the result of antibody-mediated hypersensitivity. The primary immune mediator is thought to be IgM immune complexes, as evidenced by the timing of onset prior to IgG development and the reduced occurrence over time. IgE positive test results have not been associated with hypersensitivity in any of the subjects thus far, and the majority of subjects have been safely rechallenged with rAvPAL-PEG following reactions. IgM immune complexes are known to be efficient activators of the classical complement pathway and can lead to the accumulation of complement component anaphylatoxins (C3a, C4a, C5a) that can induce hypersensitivity symptoms. Although IgG immune complexes can also activate the classical complement pathway, they do so with less efficiency than IgM. This is due, in part, to the requirement for multiple Fc regions in close proximity to activate the complement cascade, meaning that multiple monomeric IgG Abs are required to bind, whereas only one pentameric IgM Ab is needed to bind to activate complement. Also, in the case of rAvPAL-PEG, binding of anti-PAL IgG antibodies is likely compromised due to epitope masking by the PEGylation, which may reduce IgG-mediated complement activation *in vivo*. This complex dynamic between combined isotype-specific Ab responses and epitope accessibility is thought to be a major factor dictating the need for an induction and titration dose regimen in the treatment of rAvPAL-PEG to be implemented in this study.


**Table 9.1.1.2.1: Dosing Instructions in Response to Hypersensitivity Adverse Events** 

| | | Action | with Study | Drug | | |
|---|---|---|---|---|---|---|
| <u>NCI-</u><br><u>CTCAE</u><br><u>Grade<sup>a</sup></u> | Related to<br>Study Drug | <u>Maintain<sup>b</sup></u> | Reduce <sup>c</sup> | <u>Interrupt<sup>c</sup></u> | Individual<br>Stopping<br>Criteria | HRV<br>Assessment <sup>e</sup> |
| <u>1</u> | Yes or No | <u>X</u> | (X)<br>Optional | ( <u>X)</u><br>Optional | | Investigator<br>discretion |
| <u>2</u> | Yes or No | <u>X</u> | (X)<br>Optional | (X)<br>Optional | | Investigator<br>discretion |
| <u>3</u> | <u>No</u> | <u>X</u> | (X)<br>Optional | (X)<br>Optional | | Investigator<br>discretion |
| <u>3</u> | Yes | <u>X</u> | (X)<br>Optional | (X)<br>Optional | | Yes |
| and is suspected to meet Brown's criteria for severe | Yes | | | | X<br>Consult with<br>sponsor<br>medical<br>monitor | Yes |
| 4 <sup>d</sup> | Yes or No | | | | X<br>Consult with<br>sponsor<br>medical<br>monitor | Yes |

- AE, adverse event; CTCAE, Common Terminology Criteria for Adverse Events, version 4.03; HRV, Hypersensitivity Reaction Visit; NCI, National Cancer Institute.
- b NCI-CTCAE grade determination is performed by the investigator and may be done either via telephone or clinic visit.
- The investigator will instruct the subject to maintain the rAvPAL-PEG dose at the time of AE onset until improvement to grade 1 or resolution (per investigator assessment in the clinic or via telephone).
- d The rAvPAL-PEG dose may be reduced or interrupted if necessary per investigator determination.
- <sup>c</sup> If a subject has an NCI-CTCAE grade ≥ 3 hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor, the subject may be permanently discontinued from study drug.

|----------|------------|----------|

If the investigator determines that the NCI-CTCAE grade ≥ 3 hypersensitivity AE is related to administration with rAvPAL-PEG, the subject will be asked to return to the clinic within 24 hours of event onset for evaluation, including laboratory tests (chemistry, hematology, urinalysis, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE [sampling must be performed ≥8 hours after event onset and before the next dose of study drug], urine albumin/creatinine ratio, urinary N-methyl histamine, CRP, C3, C4, and tryptase).




Table 9.1.2.1: Brown's Severity Criteria

| Brown's Criteria for Hypersensitivity Reactions | <u>Definition</u> |
|---|---|
| Mild (1) skin and subcutaneous tissue | Generalized erythema, urticaria, periorbital edema, or angioedema |
| Moderate (2) features suggested respiratory, cardiovascular, or gastrointestinal involvement | Dyspnea, stridor, wheeze, nausea, vomiting, dizziness (pre-syncope), diaphoresis, chest or throat tightness, or abdominal pain |
| Severe (3) hypoxia or neurologic compromise | Cyanosis or SpO <sub>2</sub> ≤ 92% at any stage, hypotension (SBP < 90 mm Hg in adults), confusion, collapse, loss of consciousness, or incontinence |




# Vial and syringe dose to prefilled syringe dose conversion table:

| <u>Daily Dose</u><br>(mg)<br><u>Range</u> | Daily Dose<br>(mg)<br>Round To <sup>a</sup> | # of 2.5mg Prefilled Syringe Needed | # of 10mg Prefilled Syringe Needed | # of 20mg Prefilled Syringe Needed |
|---|---|---|---|---|
| <u>0 – 3.7</u> | <u>2.5</u> | <u>1</u> | <u>0</u> | <u>0</u> |
| <u>3.8 – 6.2</u> | <u>5</u> | <u>2</u> | == | == |
| 6.3 - 8.7 | <u>7.5</u> | <u>3</u> | == | == |
| 8.8 – 11.2 | <u>10</u> | = | <u>1</u> | = |
| <u>11.3 – 13.7</u> | <u>12.5</u> | <u>1</u> | <u>1</u> | == |
| 13.8 - 16.2 | <u>15</u> | <u>2</u> | <u>1</u> | = |
| <u>16.3 – 18.7</u> | <u>17.5</u> | <u>3</u> | <u>1</u> | = |
| 18.8 - 21.2 | <u>20</u> | = | II | <u>1</u> |
| 21.3 - 23.7 | <u>22.5</u> | <u>1</u> | = | <u>1</u> |
| 23.8 - 26.2 | <u>25</u> | <u>2</u> | II | <u>1</u> |
| 26.3 - 28.7 | <u>27.5</u> | <u>3</u> | = | <u>1</u> |
| <u>28.8 – 31.2</u> | <u>30</u> | = | <u>1</u> | <u>1</u> |
| <u>31.3 – 33.7</u> | <u>32.5</u> | <u>1</u> | <u>1</u> | <u>1</u> |
| 33.8 – 36.2 | <u>35</u> | <u>2</u> | <u>1</u> | <u>1</u> |
| <u>36.3 – 38.7</u> | <u>37.5</u> | <u>3</u> | <u>1</u> | <u>1</u> |
| 38.8 – 41.2 | <u>40</u> | = | = | <u>2</u> |
| 41.3 – 44.9 | <u>42.5</u> | <u>1</u> | = | 2 |
| <u>45 – 54.9</u> | <u>50</u> | = | <u>1</u> | <u>2</u> |
| <u>55 – 64.9</u> | <u>60</u> | = | = | <u>3</u> |
| <u>65 – 74.9</u> | <u>70</u> | = | <u>1</u> | 3 |
| <u>75 – 84.9</u> | <u>80</u> | = | Ξ | <u>4</u> |




| Daily Dose<br>(mg)<br>Range | <u>Daily Dose</u><br>(mg)<br><u>Round To<sup>a</sup></u> | # of 2.5mg Prefilled Syringe Needed | # of 10mg<br>Prefilled<br>Syringe Needed | # of 20mg<br>Prefilled<br>Syringe Needed |
|---|---|---|---|---|
| <u>85 – 94.9</u> | <u>90</u> | = | <u>1</u> | 4 |
| <u>95 – 104.9</u> | <u>100</u> | == | = | <u>5</u> |
| <u>105 – 114.9</u> | <u>110</u> | = | 1 | <u>5</u> |
| <u>115 – 124.9</u> | 120 | == | = | <u>6</u> |
| <u>125 – 134.9</u> | <u>130</u> | == | 1 | <u>6</u> |
| <u>135 – 144.9</u> | <u>140</u> | == | = | 7 |
| <u>145 – 154.9</u> | <u>150</u> | = | <u>1</u> | 7 |

<sup>&</sup>lt;sup>a</sup> For < 45 mg/day, round to nearest 2.5 mg; for  $\ge 45$  mg/day, round to nearest 10 mg.



# CLINICAL STUDY PROTOCOL

Study Title: Long-term Extension of a Phase 2, Open-Label, Dose-Finding

Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with

**PKU** 

Protocol Number: PAL-003

Investigational Product: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis

phenylalanine ammonia lyase)

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria (PKU)

Sponsor: BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Development Phase: Phase 2

Sponsor's Responsible Medical

Monitor:

, MD

, Clinical Sciences

BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Duration: Up to 102 months or until study is terminated

Dose: 0.001 to a maximum weekly dose of 5.0 mg/kg or 375 mg/week

Date of Original Protocol:

October 08, 2008

Date of Amendment 1:

February 09, 2009

Date of Amendment 2:

October 30, 2009

May 04, 2011

Date of Amendment 4:

June 7, 2012

Date of Amendment 5: February 28, 2014

Date of Amendment 6: October 30, 2014

Date of Amendment 7: December 16, 2015


May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

Amendment 7: 16 December 2015

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.



### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Amendment: 3

Date: 16 December 2015

### RATIONALE AND SUMMARY OF CHANGES

This section provides a numbered list of all significant changes and supporting rationale.

- 1. Collection of skin reaction data is being added to aid in assessment of skin reaction adverse events (AEs). The Skin Reaction electronic Case Report Form (eCRF) should be completed for skin reactions that last 14 days or longer. Photographs of the skin reactions may also be collected.
- 2. Additional information about subjects who are trying to conceive, are pregnant, and/or breastfeed during the study has been added. Subjects must stop study drug administration if trying to conceive, are pregnant, and/or are breastfeeding. Because of the long-term nature of this study, subjects may re-start study drug following birth and cessation of breastfeeding (if applicable) per the investigator and the sponsor. Information regarding contraception use has also been added.
- 3. The inclusion criterion regarding contraception use for subjects who are sexually active has been revised. Subjects must now use two acceptable methods of contraception while participating in the study to align with the contraception requirements in the Phase 3 studies.
- 4. The study duration has been extended from 98 months to 102 months.
- 5. The AE reporting period has been clarified; nonserious AEs and serious AEs (SAEs) should continue to be reported through 4 weeks after the last dose of study drug or the Study Completion Visit/Early Termination Visit, whichever occurs last.
- 6. Minor changes have been made to improve clarity and consistency.

In addition, the Schedule of Events and Section 12 have been updated to reflect the changes in this amendment. Refer to Section 24 for a summary of the amendment revisions.

### 2 SYNOPSIS

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

#### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


**STUDY SITES**: Approximately 20 centers in the United States

**PHASE OF DEVELOPMENT:** Phase 2

# STUDY RATIONALE:

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data were collected for subjects who have already achieved Phe reduction to within the protocol-defined target range. This substudy has been completed as of 20 December 2013.

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

# **OBJECTIVES:**

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

 To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

#### STUDY DESIGN AND PLAN:

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study. Subjects' doses will not exceed 375 mg/week.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the sponsor's medical monitor. The first dose will be administered in the clinic, and the subject must be observed for 30 minutes following administration. Additionally, subjects will be given two epinephrine injectors and will be instructed to carry one epinephrine injector with them at all times. A follow-up telephone call will be made to the subject to monitor

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self-administration. Additional training will be provided to subjects and demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (60-600  $\mu$ mol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator or Sponsor.
- The subject has completed the study through the Month 98 visit.
- The study is terminated.

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

• The study drug receives marketing authorization.

Because the risks of taking rAvPAL-PEG during pregnancy and breastfeeding are unknown, subjects cannot take rAvPAL-PEG if they are trying to conceive, are pregnant, or are breastfeeding. Male subjects who are planning to impregnate a female partner and female subjects who are trying to become pregnant during the study will be discontinued immediately from study drug. Male subjects who have impregnated a female partner may re-start study drug after conception but must return to the study-required contraception use, which must include one barrier method. Subjects who remain in the study after discontinuation of study drug due to pregnancy may re-introduce rAvPAL-PEG dosing after the birth has been reported (or termination of the pregnancy) and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to conceive. Re-starting rAvPAL-PEG dosing must be per investigator and sponsor agreement based on an assessment of the known risks and potential benefits while taking BMN 165. Female subjects must return to the study-required contraception use, which must include one barrier method, immediately after the birth (or termination of the pregnancy).

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

### PAL -003 Substudy

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed. This substudy has been completed as of 20 December 2013.

### **Dose Modifications**:

# Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| Anabaena variabilis phenylalanine ammonia lyase) NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows.

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first
  modified dose administration. Subjects who increase their dose frequency do not need to be
  observed following injection of study drug if the increase in frequency does not increase the
  overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

# Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be adjusted.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| Anabaena variabilis phenylalanine ammonia lyase) NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

### Safety Assessment Criteria:

### **Response to Hypersensitivity Adverse Events**

Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. NSAIDs should be given with food and may be omitted if not tolerated.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality. Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

### **Individual Stopping Criteria**

Subjects who have an NCI CTCAE grade  $\geq 3$  hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.

# **Dosing in Response to Hypersensitivity Adverse Events**

Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG.

Once an AE (other than anaphylaxis) improves to grade 1 or resolves, study drug dose may be increased, maintained, or reduced. If dosing has been interrupted due to an AE (other than anaphylaxis) and the investigator determines it is safe for the subject to resume dosing, the first dose after improvement of the AE should be performed in the clinic. The subject must be observed for 30 minutes following administration due to restarting dosing. The subject may be advised to premedicate with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. NSAIDs should be given with food and may be omitted if not tolerated.

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

# Response to Anaphylaxis

If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and tryptase (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then be made whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose level.

For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equipment for emergency resuscitation (including epinephrine) within easy access. The subject must be observed for 30 minutes following administration due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated.

# **Stopping Criteria:**

If an NCI-CTCAE grade ≥3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening or required treatment to prevent a life-threatening event:

- Cyanosis or  $SpO_2 \le 92\%$
- Hypotension with SBP < 90 mm Hg (adults)
- Neurologic alteration: loss of consciousness, collapse, incontinence

# **NUMBER OF SUBJECTS PLANNED:**

Up to 100 subjects.

## DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

|----------|------------|---------|
|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

- Must have completed participation in a previous rAvPAL-PEG study.
- Willing and able to provide written, signed informed consent, or, in the case of participants
  under the age of 18, provide written assent (if required) and written informed consent by a
  parent or legal guardian, after the nature of the study has been explained, and prior to any
  research-related procedures.
- Willing and able to comply with all study procedures.
- Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- Sexually active subjects must be willing to use two acceptable methods of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
- Maintained a stable diet.
- In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the sponsor's

|----------|------------|---------|
|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

medical monitor. However, subjects who discontinued from study drug early due to a reaction are not eligible to enroll into this study.

- Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- Concurrent disease or condition that would interfere with study participation or safety
  (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal,
  hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic,
  or psychiatric disease).
- Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- Known hypersensitivity to rAvPAL-PEG necessitating early termination from a previous rAvPAL-PEG study or known hypersensitivity to any of its excipients.
- Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- Creatinine > 1.5 times the upper limit of normal.

# INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self-administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing  $1.5 \pm 0.2$  mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with  $1.5 \pm 0.2$  mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

Or:

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PEG per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

Or:

|---|---|---|
| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
| BioMarin Pharmaceutical Inc. | Referring to Part of the | <b>AUTHORITY USE</b> |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |

NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase)

NAME OF ACTIVE INGREDIENT:

phenylalanine ammonia lyase

Volume: Page: Reference:

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be eligible to transition from vial and syringe to prefilled syringe dosing. Additionally, regular refresher training on use of prefilled syringe will be provided in study clinic every 24 weeks, and more often as needed.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL-PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

# **Fixed Dosing**

Subjects who have demonstrated efficacy (ie, blood Phe within the target range of  $60-600 \mu mol/L$  for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week).

# **DURATION OF TREATMENT:**

Up to 102 months.

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

# CRITERIA FOR EVALUATION:

# Efficacy:

Blood Phe concentrations will be measured.

|----------|------------|---------|
|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

# Immunogenicity:

The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-PEG neutralizing antibodies, anti-rAvPAL IgE, and anti-PEG-PAL IgE) will be assessed.

# **Safety**:

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs, ECG results, X-ray results, and laboratory test results.

# **Pharmacokinetic**:

Plasma concentrations of rAvPAL-PEG will be measured for subjects participating in the Substudy.

# **STATISTICAL METHODS:**

# Sample Size:

Subjects who participated in a previous rAvPAL-PEG study may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

# **Safety Analysis:**

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by-subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided.

|----------|------------|---------|
|----------|------------|---------|

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY USE |
| 105 Digital Drive | Dossier: | ONLY: |
| Novato, CA 94949 | | |
| | Volume: | |
| rAvPAL-PEG (PEGylated recombinant | Reference: | |
| Anabaena variabilis phenylalanine ammonia | | |
| lyase) | | |
| NAME OF ACTIVE INGREDIENT: | | |
| phenylalanine ammonia lyase | | |

Descriptive statistics for vital signs, physical examination results, ECG results, X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

# **Efficacy Analysis**:

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the Statistical Analysis Plan [SAP]) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

### **Exploratory Analysis:**

Details regarding exploratory analyses will be provided in the SAP.

# **Substudy Analysis:**

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

# Pharmacokinetic Analysis:

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F).

| <b>B</b> OMARIN | B | 0 | M | A | R | IN |
|-----------------|---|---|---|---|---|----|
|-----------------|---|---|---|---|---|----|


# 3 TABLE OF CONTENTS

| 1 | TIT | LE PAG | 6E | 1 |
|---|---|---|---|---|
| 2 | SYN | NOPSIS | | 3 |
| 3 | TAE | BLE OF | CONTENTS | 15 |
| 4 | LIS | T OF AI | BBREVIATIONS AND DEFINITIONS OF TERMS | 19 |
| 5 | ETH | HCS | | 23 |
| | 5.1 | Institut | tional Review Board or Ethics Committee | 23 |
| | 5.2 | Ethical | l Conduct of Study | 23 |
| | 5.3 | Subjec | et Information and Informed Consent | 24 |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 25 |
| 7 | INT | RODUC | CTION | 26 |
| | 7.1 | Noncli | inical Studies | 26 |
| | 7.2 | Previo | us Clinical Studies | 27 |
| | | 7.2.1 | Phase 1 Study, PAL-001 | 28 |
| | | 7.2.2 | Phase 2 Studies PAL-002, PAL-004, and 165-205 | 28 |
| | 7.3 | Study | Rationale | 32 |
| | 7.4 | Summ | ary of Overall Risks and Benefits | 33 |
| | | 7.4.1 | Toxicity Due to Exposure to Polyethylene Glycol (PEG) | 33 |
| | | 7.4.2 | Immunologic Response | 34 |
| | | 7.4.3 | Management of Hypersensitivity Reactions | 35 |
| 8 | STU | JDY OB | JECTIVES | 37 |
| 9 | INVESTIGATIONAL PLAN | | 38 | |
| | 9.1 | Overal | ll Study Design and Plan | 38 |
| | | 9.1.1 | Response to Hypersensitivity Adverse Events | 45 |
| | | 9.1.2 | Study Stopping Criteria | 47 |
| | | 9.1.3 | Dose Modifications | 48 |
| | 9.2 | Discus | ssion of Study Design, Including Choice of Control Group | 49 |
| | 9.3 | Selecti | ion of Study Population | 49 |
| | | 9.3.1 | Inclusion Criteria | 49 |
| | | 9.3.2 | Exclusion Criteria | 50 |

| BIC | MA | RIN | PAL-003 A7 | Page 16 |
|---|---|---|---|---|
| | 9.3.3 | Removal | of Subjects from Treatment or Assessment | 51 |
| | 9.3.4 | | entification and Replacement of Subjects. | |
| 9.4 | | | | |
| 2.1 | 9.4.1 | | s Administered | |
| | 9.4.2 | | f Investigational Product (IP) | |
| | 9.4.3 | | · | |
| | 9.4.4 | _ | for Administration | |
| | 9.4.5 | | f Assigning Subjects to Treatment Groups | |
| | 9.4.6 | | of Doses Used in the Study | |
| | 9.4.7 | | | |
| | 9.4.8 | | Concomitant Medications | |
| | 9.4.9 | | Compliance | |
| | 9.4.10 | | ruption and Missed Doses | |
| 9.5 | Investig | | oduct Accountability | |
| | 9.5.1 | | d Disposition of Clinical Supplies | |
| 9.6 | Dietary | | rotocol Restrictions | |
| 9.7 | _ | | y Variables | |
| | 9.7.1 | Efficacy a | nd Safety Measurements Assessed | 62 |
| | 9.7.2 | Efficacy V | /ariable | 64 |
| | 9.7.3 | Pharmaco | kinetic Variables | 64 |
| | 9.7.4 | Explorato | ry Efficacy Variable | 65 |
| | 9.7.5 | Safety Va | riables | 65 |
| | 9.7.6 | Clinical L | aboratory Assessments | 65 |
| 10 REP | ORTING | G ADVERS | SE EVENTS | 68 |
| 10.1 | Adverse | e Events | | 68 |
| 10.2 | Serious | Adverse E | vents | 70 |
| 10.3 | Pregnar | ncy | | 72 |
| 10.4 | Urgent | Safety Mea | isures | 72 |
| 10.5 | BioMar | rin Pharmac | covigilance Contact Information | 73 |
| 11 APP | R OPRIA | TENESS ( | OF MEASUREMENTS | 72 |

| | OMARIN | PAL-003 A / | Page 17 |
|---|---|---|---|
| | 11.1 Safety and Pharma | cokinetics | 72 |
| 12 | - | S | |
| - | | | |
| | | eek 1) | |
| | | elephone Visit | |
| | | Visits | |
| | • | Visits (Week 4, 8, 12, etc) | |
| | • | Visits (Week 12, 24, 36, etc) | |
| | | led Hypersensitivity Reaction Visit | |
| | | /Early Termination Visit | |
| 13 | | URANCE | |
| | | ODS AND DETERMINATION OF SAMPI | |
| | 14.1 Statistical and Ana | ılytical Plans | 81 |
| | 14.3 Pharmacokinetic A | Analysis | 81 |
| | 14.3.1 Pharmaco | kinetic Substudy Analysis | 82 |
| | 14.5 Determination of S | Sample Size | 82 |
| | 14.6 Handling of Missi | ng Data | 82 |
| | 14.7 Interim Analyses | | 83 |
| | 14.8 Changes in the Co | nduct of the Study or Planned Analyses | 83 |
| 15 | DATA MONITORING | COMMITTEE (DMC) | 84 |
| 16 | COMPENSATION, INS | SURANCE, AND INDEMNITY | 85 |
| 17 | CASE REPORT FORM | S AND SOURCE DOCUMENTS | 86 |
| 18 | STUDY MONITORING | G AND AUDITING | 87 |
| 19 | RETENTION OF RECO | ORDS | 88 |
| 20 | USE OF INFORMATIO | ON AND PUBLICATION | 80 |

| <b>B</b> IOMARIN | PAL-003 A7 | Page 18 |
|---|---|---|
| 21 REFERENCES | | 90 |
| 22 INVESTIGATOR RESE | PONSIBILITIES | 92 |
| 22.1 Conduct of Study a | and Protection of Human Subjects | 92 |
| 24 PROTOCOL AMENDM | MENT TEXT REVISIONS | 94 |
| LIST OF TABLES | | |
| Table 9.1.1: Schedule of Ev | vents | 41 |
| Table 9.1.2: PK Substudy D | Oosing Regimens | 44 |
| Table 9.1.1.2.1: Dosing Inst | tructions in Response to Hypersensitivity | Adverse Events46 |
| Table 9.1.2.1: Brown's Sev | erity Criteria | 48 |
| Table 9.4.2.1.1: Prefilled Sy | yringe Volume, Concentration, and Dose. | 55 |
| Table 9.4.2.1.2: Conversion | from Vial and Syringe Dose to Prefilled | Syringe Dose56 |
| Table 9.4.4.1: Fixed Doses | for Subjects on Weight-Based Dose Regin | men58 |
| Table 9.7.1.1: Summary of | Laboratory Assessments | 63 |
| Table 9.7.6.1: Clinical Laboratory | oratory Tests | 67 |




# 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# **Abbreviations**

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

AUC<sub>0-7 davs</sub> area under the plasma concentration-time curve from time zero on Day 1

to Day 8

BUN blood urea nitrogen
°C degree Celsius
C<sub>3</sub> complement 3
C<sub>4</sub> complement 4

CBC complete blood count

CD Compact disk

CFR Code of Federal Regulations
CH50 total hemolytic complement
C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form
CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure

DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up g gram

GCP Good Clinical Practice

|----------|------------|---------|
|----------|------------|---------|

GGT gamma-glutamyltransferase

GI gastrointestinal

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

ID identification

IgEimmunoglobulin EIgGimmunoglobulin GIgMimmunoglobulin MIPinvestigational productIRBInstitutional Review Board

IV intravenous kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

NAb neutralizing antibodies

NCI National Cancer Institute

NIAID/FAAN National Institute of Allergy and Infectious Disease/Food Allergy and

Anaphylaxis Network

NOAEL no observable adverse effect level

NSAID non-steroidal anti-inflammatory medication

OTC over the counter

PAH phenylalanine hydroxylase PAL phenylalanine ammonia lyase

PEG polyethylene glycol

Phe phenylalanine

PI Principal Investigator
PK pharmacokinetics
PKU phenylketonuria

rAvPAL-PEG recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG

RBC red blood cell
|----------|------------|---------|
|----------|------------|---------|

SAE serious adverse event
SAP Statistical Analysis Plan
SBP systolic blood pressure

SC subcutaneous

SD standard deviation SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase SGPT serum glutamic pyruvate transaminase

US United States
WBC white blood cell

|----------|------------|---------|
|----------|------------|---------|

## Definition of Terms:

Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.

| <b>B</b> OMARIN | PAL-003 A7 | Page 23 |
|-----------------|------------|---------|
|-----------------|------------|---------|

#### 5 ETHICS

#### 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

## 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will



provide written, informed consent before any study-related tests or evaluations are performed.

## 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR Part 50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



#### 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Pharmacovigilance Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations and urinalysis. Pharmacokinetic (PK) analysis will be performed by BioMarin.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.

|----------|------------|---------|
|----------|------------|---------|

#### 7 INTRODUCTION

A comprehensive review of PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

## 7.1 Nonclinical Studies

The nonclinical program for rAvPAL-PEG has characterized the pharmacology, pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC route of administration. Pharmacology was assessed in the BTBR  $Pah^{\rm enu2}$  (ENU2) mouse model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to 2000  $\mu$ M) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to male ENU2 mice, plasma Phe concentrations decreased from approximately 2000  $\mu$ M to < 200  $\mu$ M after 2 dose administrations. An attenuated reduction of blood Phe was seen between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe < 200  $\mu$ M over the entire week, which continued for a total of 15 weeks.

In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a 2-4 week dose interruption and an 11-week dose interruption. Following both dose interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A similar interim attenuated response was observed with the longer dose interruption of approximately 11 weeks. In both of these assessments, no safety issues were noted upon re-starting dosing with rAvPAL-PEG (Lapis, 2007, ASHG 57th Annual Meeting).

Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No respiratory or central nervous system (CNS) effects were seen with SC administration of rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV effects of rAvPAL-PEG administered subcutaneously.

Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats and cynomolgus monkeys. The elimination half-life ( $t_{1/2}$ ) values of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and 44 hours, respectively,

| BIOM | AR | N. |
|------|----|----|
|------|----|----|


and exhibited modest area under the plasma concentration-time curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the  $t_{1/2}$  was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum observed plasma concentration ( $C_{max}$ ), along with a long  $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) the AUC and the  $C_{max}$  are roughly linearly proportional.

Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given  $\geq 3$  mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey.

#### 7.2 Previous Clinical Studies

The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002, Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience from this ongoing study and the other ongoing Phase 2 studies, PAL-002 and PAL-004.



# 7.2.1 Phase 1 Study, PAL-001

The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations.

The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 µmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG.

Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows:

- rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg.
- For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level for these 5 subjects was 1113 µmol/L.
- Overall, no clinically significant reductions in blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, 0.01, and 0.03 mg/kg.
- For subjects who were administered rAvPAL-PEG at the 3 higher dose levels (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration levels, the calculated PK parameters were a mean T<sub>max</sub> of 89-106 hours, a t<sub>1/2</sub> of 46-120 hours, and an AUC<sub>0-t</sub>, and C<sub>max</sub> that were proportional with dose. Drug exposure was slightly increased with increased dose.

## 7.2.2 Phase 2 Studies PAL-002, PAL-004, and 165-205

Based on results from the Phase 1, single-dose study, the Phase 2 studies have been designed to evaluate rAvPAL-PEG at various doses and dosing regimens to safely achieve and maintain blood Phe reductions in subjects with PKU. Currently, there are three ongoing Phase 2 studies (PAL-002, PAL-004, 165-205); an overview of each study is presented in Section 7.2.2.1 (PAL-002), Section 7.2.2.2 (PAL-004), and Section 7.2.2.3 (165-205).

|----------|------------|---------|
|----------|------------|---------|

### 7.2.2.1 Study PAL-002

Study PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria) was initiated in September 2009 and has completed enrollment. As of 10 September 2012, 40 subjects have been enrolled and 37 have completed the study. PAL-002 enrolled 11 previously exposed subjects from the single-dose study, PAL-001, and 29 subjects who were naïve to rAvPAL-PEG. Thirty-three of the 37 subjects who completed PAL-002 enrolled into this open-label extension study (PAL-003). Two subjects discontinued from the study due to lost to follow-up, relocation, or other reasons, and 1 subject discontinued from the study due to an AE (skin reaction).

The primary objective of this study was to evaluate the effect of multiple doses of rAvPAL-PEG (ranging from 0.001 mg/kg/week to 1.0 mg/kg/week) on blood Phe concentrations in subjects with PKU with up to 16 weeks of treatment. The secondary objectives of the study were to evaluate the safety and tolerability of SC injections of multiple doses of rAvPAL-PEG, to evaluate the immune response to rAvPAL-PEG, and to evaluate the PK profile of rAvPAL-PEG in subjects with PKU.

The PAL-002 study design consists of two parts. In Part 1, rAvPAL-PEG was administered as a once weekly fixed, low-dose induction regimen for 8 weeks. In Part 2, the rAvPAL-PEG dose was titrated upwards; subjects received adjustable dose increases for up to 8 weeks to achieve a target blood Phe concentration of 600 µmol/L. The doses and dosing schedules were revised with a series of protocol amendments to incorporate the information gained during conduct of this early, open-label, multiple-dose study.

A wide range of doses was planned for the PAL-002 study, beginning with doses as low as 0.001 mg/kg/week. However, no substantial reductions in blood Phe level were observed in the majority of subjects who were administered rAvPAL-PEG in the initial four cohorts at doses of 0.001, 0.003, 0.01, and 0.03 mg/kg administered once per week. The absence of appreciable Phe reduction after 16 weeks of treatment in this range of doses led to a decision to amend the study protocol to include a cohort with a higher starting dose of 0.1 mg/kg/week, which had been previously shown to decrease blood Phe levels to approximately  $600 \text{ }\mu\text{mol/L}$  in the single-dose, Phase 1 study (PAL-001). After the first 2 weeks of dosing at 0.1 mg/kg/week, transient Phe reduction was observed in this subset of subjects. However, this dosing regimen was accompanied by mild to moderate hypersensitivity reactions primarily after the second weekly dose, suggesting that additional exploration of dosing regimens would be required.


| <b>B</b> OMARIN | PAL-003 A7 |
|-----------------|------------|
|-----------------|------------|

In summary, preliminary results from PAL-002 demonstrated that doses below 0.1 g/kg administered once per week were not effective in reducing Phe levels. While transient reduction of Phe was apparent at doses of at least 0.1 mg/kg given once per week, this dose regimen was associated with a high incidence of systemic hypersensitivity reactions, typically following the second weekly dose. Further escalation above this dose of 0.1 mg/kg/week would be required to sustain the effect on Phe levels over time. Increased doses would require spreading dose administration over several days per week, as once-weekly administration of higher doses would not be practical due to the large volume of study drug. Therefore, additional dosing regimens would need to be explored in a subsequent study (PAL-004).

Once subjects completed Study PAL-002, they were eligible to enroll into this open-label extension study, PAL-003 to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

## 7.2.2.2 Study PAL-004

PAL-004 (An Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Dose Levels of rAvPAL-PEG Administered Daily in Subjects With Phenylketonuria) was initiated in April 2011 and has completed enrollment. As of 10 September 2012, 16 subjects have been enrolled, 15 subjects have completed the study, and 15 subjects have enrolled into this study (PAL-003). One subject withdrew consent from continued participation prior to study completion. All subjects enrolled in this study were naïve to rAvPAL-PEG exposure.

The objective of this study was to determine if daily administration (defined as 5days/week) of rAvPAL-PEG at dose levels of 0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day was safe and effective in reducing and maintaining blood Phe concentrations to 600 µmol/L in subjects with PKU. The starting dose was 0.4 mg/kg, administered 5 days/week. A total of 12 subjects were added in sequence and were started on doses of 0.4, 0.2, 0.1, 0.06 mg, or 0.001/kg/day based on incoming safety data. Overall, subjects in PAL-004 who initiated treatment at higher daily doses of 0.1 to 0.4 mg/kg/day achieved immediate and substantial reduction of blood Phe levels, but dosing had to be temporarily reduced or interrupted due to the onset of systemic hypersensitivity reactions at approximately Day 10 of dosing. Phe reductions did not persist in the setting of temporary dose reduction or interruption, but Phe levels generally improved if higher dose levels were reinstated.

To prevent the onset of hypersensitivity reactions that were temporally associated with the onset of anti-drug IgM responses, an additional dosing strategy was assessed in PAL-004;

| BIO | M | A | R | IN | 00 |
|-----|---|---|---|----|----|
|-----|---|---|---|----|----|


4 subjects initiated dosing at a low dose of 0.001mg/kg/day or 0.06mg/kg/day for 5 consecutive days and then dosing was suspended for 2 weeks. Dosing was restarted on Day 21 at the initial dose followed by dose titration to target Phe levels. Subjects administered this dosing regimen had similar efficacy, but the incidence of hypersensitivity reactions appeared to be similar to that of subjects who did not have the planned dose interruption, suggesting little advantage with this alternate induction regimen.

Experience from PAL-004 indicated that initiating daily rAvPAL-PEG dosing with relatively high daily doses was not sustainable due to the onset of hypersensitivity reactions that occurred approximately 9 to 12 days after the start of administration, nor was the alternate dosing regimen (2 week drug holiday) well tolerated or effective in Phe reduction. In addition, the daily treatment regimen did not reduce the time to achieve target blood Phe levels seen in previous studies. This study indicated that to improve tolerability, rAvPAL-PEG should be initiated with an induction period at doses substantially lower than 0.4mg/kg, followed by upward dose titration toward target Phe levels.

Once subjects completed Study PAL-004, they were eligible to enroll into this open-label extension study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

## 7.2.2.3 Study 165-205

Study 165-205 (A Phase 2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate Safety, Efficacy, and Tolerability of Subcutaneously Administered rAvPAL-PEG in Subjects With PKU for 24 Weeks) was initiated in May 2012. Data from ongoing Studies PAL-002, PAL-004, and PAL-003 suggested that a 4-week treatment course with weekly dosing at a fixed low dose (induction), followed by a weekly 2-fold, upward titration of rAvPAL-PEG to approximately 10-fold higher than the initiation dose (maximum of 375 mg/week) is effective and well tolerated. The objective of this study was to further assess this dosing regimen. Two rAvPAL-PEG dosing regimens were to be explored in this study: weekly low-dose induction (2.5 mg/week for 4 to 8 weeks), followed by a period of upward dose titration towards a target Phe level (600 µmol/L) followed by maintenance dosing at that level through the 24 week study duration (Group 1). The other dosing regimen planned for this study (Group 2) involved administration of a single bolus dose of 8 mg, followed by a treatment holiday of at least 3 weeks duration followed by resumption and escalation of study drug administration following a pattern similar to that employed in Group 1. A total of 24 subjects were enrolled into 165-205. In addition to confirming an effective, well-tolerated dose regimen, this study incorporated non-weight-based dosing, starting with dose

|----------|------------|---------|
|----------|------------|---------|

administration once per week at a low dose (2.5mg) with gradual escalation and conversion of dose administration to 5x/week dosing for chronic maintenance therapy.

Once subjects have completed Study 165-205, they are eligible to enroll into this study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week, or into the Phase 3 study, 165-302.

## 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH. Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan® is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. rAvPAL-PEG is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an

| <b>B</b> IOMARIN | PAL-003 A7 | Page 33 |
|------------------|------------|---------|
|------------------|------------|---------|

exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

This study is an extension of previous rAvPAL-PEG Phase 2 studies. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

### 7.4 Summary of Overall Risks and Benefits

It is not expected that data from previous rAvPAL-PEG studies will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

## 7.4.1 Toxicity Due to Exposure to Polyethylene Glycol (PEG)

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg rAvPAL-PEG SC. In rats, both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1).

| SIN. | RI | MA | 0 | B |
|------|----|----|---|---|
|------|----|----|---|---|


In this study, subjects will be monitored closely with urine examinations and blood chemistries to follow kidney function.

## 7.4.2 Immunologic Response

The active drug substance in rAvPAL-PEG is a bacterial protein and elicits immune recognition and subsequent antibody responses. Antibody epitopes on the protein are expected to be rendered at least partially inaccessible by the extensive PEGylation on the drug (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in reducing anti-rAvPAL antibody titers in the mouse model but does not eliminate antibody formation. Although PEGylation of rAvPAL likely reduces the antigenicity of the molecule, 100% of individuals exposed to rAvPAL-PEG develop antibodies against rAvPAL.

Drug-specific immune responses can range from clinical irrelevance to causing serious hypersensitivity AEs (such as anaphylaxis) and may reduce efficacy due to antibody-mediated drug clearance or antibody neutralization of enzymatic activity. Historically, PEG was thought to be nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.), (Harris, 2003, Nat.Rev.Drug Discov.); however, repeated studies have found that subcutaneous (SC) and intravenous exposure to PEG can induce anti-PEG antibodies (Harris, 2003, Nat.Rev.Drug Discov.), (Richter, 1983, Int.Arch.Allergy Appl.Immunol.). In some instances, development of such antibodies did not result in significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). However, PEG antibody responses were associated with hypersensitivity reactions to PEGylated liposomes (Judge, 2006, Mol.Ther.). Anti-PEG antibodies have also been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.).

Subjects participating in the Phase 2 clinical studies have been monitored closely for anti-drug immunogenicity (anti-rAvPAL immunoglobulin G [IgG], anti-rAvPAL IgM, anti-PEG IgM, anti-PEG IgG, neutralizing antibodies that inhibit PAL enzymatic activity, anti-rAvPAL IgE, and anti-rAvPAL-PEG IgE), complements, C-reactive protein (CRP), ESR, and complete chemistry. All subjects treated with rAvPAL-PEG in the Phase 2 clinical trials developed antibodies against the PAL protein. Anti-rAvPAL IgM antibodies were first detected within 2-3 weeks of treatment initiation and anti-rAvPAL IgG antibodies were detected within 2-3 months. The anti-rAvPAL IgG response generally peaked by 3-5 months and was sustained in all subjects. Neutralizing antibodies (NAb) capable of inhibiting enzymatic activity were detected in a minority of subjects 2-3 months after treatment initiation. The timing of the NAb response suggests these antibodies may be a component of

| <b>B</b> OMARIN | PAL-003 A7 | Page 35 |
|-----------------|------------|---------|
|-----------------|------------|---------|

the anti-rAvPAL IgG response. It is expected that the centralized location of the PAL active site, within the tetrameric structure, makes it difficult for antibodies to bind and inhibit enzymatic activity. In addition, anti-PAL antibody binding is likely sterically hindered by the extensive PEGylation. The majority of treated subjects also developed a transient anti-PEG antibody response. The anti-PEG response was comprised of IgM and IgG isotypes. In general, anti-PEG antibodies were no longer detected after 5-6 months of treatment. This type of transient antibody response is typical of T cell-independent type 2 (TI-2) responses.

The majority of immune-mediated AEs experienced in subjects treated with rAvPAL-PEG in the Phase 2 studies are believed to be the result of antibody-mediated hypersensitivity. The primary immune mediator is thought to be IgM immune complexes, as evidenced by the timing of onset prior to IgG development and the reduced occurrence over time. IgE positive test results have not been associated with hypersensitivity in any of the subjects thus far, and the majority of subjects have been safely rechallenged with rAvPAL-PEG following reactions. IgM immune complexes are known to be efficient activators of the classical complement pathway and can lead to the accumulation of complement component anaphylatoxins (C3a, C4a, C5a) that can induce hypersensitivity symptoms. Although IgG immune complexes can also activate the classical complement pathway, they do so with less efficiency than IgM. This is due, in part, to the requirement for multiple Fc regions in close proximity to activate the complement cascade, meaning that multiple monomeric IgG Abs are required to bind, whereas only one pentameric IgM Ab is needed to bind to activate complement. Also, in the case of rAvPAL-PEG, binding of anti-PAL IgG antibodies is likely compromised due to epitope masking by the PEGylation, which may reduce IgG-mediated complement activation in vivo. This complex dynamic between combined isotype-specific Ab responses and epitope accessibility is thought to be a major factor dictating the need for an induction and titration dose regimen in the treatment of rAvPAL-PEG to be implemented in this study.

## 7.4.3 Management of Hypersensitivity Reactions

Hypersensitivity reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 30 minutes post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of hypersensitivity reactions. Because of the potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection. Subject should be pre-medicated with H1 antagonist, H2

| <b>B</b> IOMARIN | PAL-003 A7 | Page 36 |
|------------------|------------|---------|
|------------------|------------|---------|

antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated. Subjects who qualify for self-administration of study drug are trained to recognize a serious hypersensitivity AEs and how to respond. Additionally, subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (Section 9.4). Refer to Section 9.1.1.3 for instructions regarding resumption of study drug following resolution of symptoms consistent with a clinical diagnosis of anaphylaxis per National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria (Sampson, 2006, J.Allergy Clin.Immunol.).

In the event of a hypersensitivity reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for immunology studies and complement testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of hypersensitivity reaction symptoms:

- Maintain the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oral or IV glucocorticoids.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. An allergy and/or immunology consultation should be sought if necessary. Detailed instructions for the management of hypersensitivity reactions are provided in the Study Reference Manual.

| <b>B</b> IOMARIN | PAL-003 A7 | Page 37 |
|------------------|------------|---------|
|------------------|------------|---------|

#### 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objective is as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.



#### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity was observed in a previous rAvPAL-PEG studies. Subjects' doses will not exceed 375 mg/week.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the sponsor's medical monitor. The first week of dosing will be administered in the clinic, and the subject must be observed for 30 minutes following administration. Subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (refer to Section 9.4). A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to clinic monthly for review with the clinical study staff.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self-administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self-administration. Additional information is provided in the Subject Self-Administration Training Materials. Additional training will be provided and demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

|----------|------------|---------|
|----------|------------|---------|

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 9.1.1 and Table 9.1.2. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator or Sponsor.
- The subject has completed the study through the Month 98 visit.
- The study is terminated.
- The study drug receives marketing authorization.

Because the risks of taking rAvPAL-PEG during pregnancy and breastfeeding are unknown, subjects cannot take rAvPAL-PEG if they are trying to conceive, are pregnant, or are breastfeeding (refer to Section 9.3.2, Exclusion Criteria). Male subjects who are planning to impregnate a female partner and female subjects who are trying to become pregnant during the study will be discontinued immediately from study drug. Male subjects who have impregnated a female partner may re-start study drug after conception but must return to the study-required contraception use (refer to Section 9.3.1, Inclusion Criteria), which must include one barrier method. Subjects who remain in the study after discontinuation of study drug due to pregnancy may re-introduce rAvPAL-PEG dosing after the birth has been reported (or termination of the pregnancy) and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to conceive. Re-starting rAvPAL-PEG dosing must be per investigator and sponsor agreement based on an assessment of the known risks and potential benefits while taking BMN 165. Female subjects must return to the



study-required contraception use (refer to Section 9.3.1), which must include one barrier method, immediately after the birth (or termination of the pregnancy).

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed (refer to Table 9.1.2).

The Schedule of Events and PK substudy collection schedules are presented below in Table 9.1.1 and Table 9.1.2.

|----------|------------|---------|
|----------|------------|---------|

**Table 9.1.1: Schedule of Events** 

| | | | Tre | eatment Perio | od <sup>b,c</sup> | | | |
|---|---|---|---|---|---|---|---|---|
| | | Week<br>1 | Weekly<br>Telephone<br>Contacts | Monthly b<br>(eg, Wk 4,<br>8, etc.) | Quarterly<br>(eg, Wk 12,<br>24, etc.) | Self-<br>Administration | Study<br>Completion/Early<br>Term. Visit | |
| Assessments and Events | Screening <sup>a</sup> | D1 | Starting at<br>Week 2 | Every 4th week; | Every 12th week. Perform in addition to monthly procedures | | 4 weeks after<br>final dose | Unsched. Hyper.<br>Reaction Visit. <sup>d</sup><br>Perform within<br>24 hours |
| Informed consent | X | | | | | | | |
| Medical history, including allergy history, and demographics | Λ | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | | X | | X | |
| Vital signs <sup>e</sup> | X | X | | X | | | X | X |
| Weight | X | | | X | | | | |
| 12-lead ECG | X | | | | | | X | |
| Clinical laboratory tests <sup>f</sup> | X | | | X | | | X | Xg |
| Complements C <sub>3</sub> and C <sub>4</sub> <sup>h</sup> | X | | | | X | | | Xg |
| Sedimentation rate | | X | | | X | | X | |
| Chest x-ray | X | | | X<br>(Week 48<br>visit only) | | | X | |
| Urine pregnancy test <sup>i</sup> | X | X | | X | | | X | |
| Adverse events <sup>j,k</sup> | X | X | X | X | | X | X | X |
| Weekly phone call to self admin<br>participants only (to assess AEs,<br>Inj site reactions, concomitant<br>medications) | | | X | | | X | | |
| Concomitant medications | X | X | X | X | | X | X | X |
| Diet query | X | X | | X | | | X | |
| 3-Day diet diary <sup>1</sup> | | | | X | | | X | |
| Serum antibodies <sup>m</sup> | | X | | | X | | X | X |

| B <b>!</b> OMARIN | PAL-003 A7 | Page 42 |
|-------------------|------------|---------|
|-------------------|------------|---------|

| | | | Tro | eatment Perio | od <sup>b,c</sup> | | | |
|---|---|---|---|---|---|---|---|---|
| | | Week<br>1 | Weekly<br>Telephone<br>Contacts | Monthly b<br>(eg, Wk 4,<br>8, etc.) | Quarterly (eg, Wk 12, 24, etc.) | Self-<br>Administration | Study<br>Completion/Early<br>Term. Visit | |
| Assessments and<br>Events | Screeninga | D 1 | Starting at<br>Week 2 | Every 4th<br>week; | Every 12th week. Perform in addition to monthly procedures | | 4 weeks after<br>final dose | Unsched. Hyper.<br>Reaction Visit. <sup>d</sup><br>Perform within<br>24 hours |
| Plasma Phe and plasma tyrosine <sup>n</sup> | X | X | | $X^{m}$ | | | X | |
| Urine albumin/creatinine ratio | | | | | | | | X |
| Urine N-methyl histamine | | | | | | | | X |
| Plasma PK sample <sup>o</sup> | | X | | | X | | X | |
| Administer study drug <sup>p</sup> | | X | | X | | X | | |
| Training (prefilled syringe) <sup>q</sup> | | | | X<br>Transition<br>to prefilled<br>syringe | X<br>Every 24<br>weeks only | | | |
| Skin biopsy (optional; affected and not affected area) | | | | | | | | X |
| Serum tryptase level <sup>r</sup> | | | | | | | | X |

AE, adverse event; C<sub>3</sub>, complement 3; C<sub>4</sub>, complement 4; CH50, total hemolytic complement; CRP, C-reactive protein; D, day; ECG, electrocardiogram; eCRF, electronic Case Report Form; ETV, Early Termination Visit; F/U, Follow-up; Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> A separate Screening visit for this study is required only if the time between completion of the previous rAvPAL-PEG study and enrollment into PAL-003 is greater than 28 days.

<sup>&</sup>lt;sup>b</sup> Monthly visits must be performed in the clinic.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Refer to Section 9.1.1 and Section 12.3.6.

<sup>&</sup>lt;sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.

|----------|------------|---------|
|----------|------------|---------|

<sup>&</sup>lt;sup>f</sup> Clinical laboratory tests to include spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis. Urine microscopy will be performed if any urinalysis results are positive for hematuria. Refer to Table 9.7.6.1.

- <sup>g</sup> Subjects who have a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade ≥ 3 hypersensitivity AE should be assessed for CRP, CH50, C1, C3, and C4 within 24 hours of the reaction.
- <sup>h</sup> Complement C3 and C4 will be collected at the Screening Visit and quarterly. Additional complement testing will be performed and as needed to resolve previous abnormal test results.
- <sup>i</sup> If positive or equivocal, perform serum pregnancy test. Also refer to Section 9.1.
- j If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm). If there is a skin reaction that lasts ≥ 14 days, the Skin Reaction eCRF should be completed. A photograph of the skin reaction may be taken by the subject or the site to help assess the event and may be collected by the sponsor.
- <sup>k</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or completion of study participation, whichever occurs last. The reporting period for nonserious AEs is from the first administration of study drug through 4 weeks after last dose or the Study Completion Visit/Early Termination Visit, whichever occurs last. The reporting period for device-related events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe.
- <sup>1</sup> It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.
- <sup>m</sup> For unscheduled hypersensitivity reaction visit, draw serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only; sampling must be performed > 8 hours after event onset and before the next dose of study drug.
- <sup>n</sup> Samples should be drawn at least 2.5 hours after a meal. At the Investigator's discretion, blood Phe may be collected more often should more frequent monitoring of blood Phe levels be clinically warranted.
- ° Sampling should be performed predose.
- <sup>p</sup> Dosing is up to 5.0 mg/kg/week or 375 mg/week, including subjects who receive more than 1 dose/week. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may be re-evaluated.
- <sup>q</sup> Initial training on the use of prefilled syringe occurs at the next monthly visit and each subsequent day after transition until (in clinic or by HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter.
- <sup>r</sup> Mandatory for subjects who have a hypersensitivity AE. Perform within 24 hours of event onset.

|----------|------------|---------|
|----------|------------|---------|

**Table 9.1.2: PK Substudy Dosing Regimens** 

| <b>Treatment Frequency</b> | Plasma PK Sampling | Example |
|---|---|---|
| Subjects who are<br>administered study drug<br>once per week | Pre-dose and every 24 hours<br>thereafter (24, 48, 72, and 96<br>hours when possible), and<br>pre-dose of the next weekly<br>dose | If dosed on Monday: Obtain PK sample pre-dose when possible – pre-dose Monday, Tuesday, Wednesday, Thursday, Friday, and pre-dose the following Monday. No further PK substudy draws. |
| Subjects who are<br>administered study drug<br>two or three times per<br>week | Pre-dose and every 24 hours<br>during the longest period<br>between doses, when<br>possible, and pre-dose of the<br>next dose. | If dosed on Monday, Thursday, and Friday: Obtain PK sample every 24 hours during the longest period between doses: Pre-dose Monday, Tuesday, Wednesday, and pre-dose Thursday. No further PK substudy draws. |
| Subjects who are administered study drug four to seven times per week. | Pre-dose and every 12 hours during the longest period between doses, when possible, then pre-dose of the next dose. | If dosed Monday through Friday: Obtain PK sample every 12 hours during the longest period between doses (Friday to Monday): pre-dose Friday, 12 hours post-dose Friday, Saturday (24 and 36 hours post dose), Sunday (48 and 60 hours post-dose), and pre-dose the following Monday. No further PK substudy draws. |



# 9.1.1 Response to Hypersensitivity Adverse Events

Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. NSAIDs should be given with food and may be omitted if not tolerated.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality (Section 9.1.1.3). Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

## 9.1.1.1 Individual Stopping Criteria

Subjects who have an NCI CTCAE grade  $\geq 3$  hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.

#### 9.1.1.2 Dosing in Response to Hypersensitivity Adverse Events

Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG. Dosing instructions are presented in Table 9.1.1.2.1 and are regardless of previous occurrence:



**Table 9.1.1.2.1: Dosing Instructions in Response to Hypersensitivity Adverse Events** 

| NCI-CTCAE | Related to | Action | with Stud | y Drug | Individual<br>Stopping | HRV |
|---|---|---|---|---|---|---|
| <b>Grade</b> <sup>a</sup> | Study Drug | Maintain <sup>b</sup> | Reducec | Interrupt <sup>c</sup> | Criteria d | Assessment <sup>e</sup> |
| 1 | Yes or No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 2 | Yes or No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 3 | No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 3 | Yes | X | (X)<br>Optional | (X)<br>Optional | | Yes |
| and is suspected to<br>meet Brown's<br>criteria for severe d | Yes | | | | X Consult with sponsor medical monitor | Yes |
| 4 <sup>d</sup> | Yes or No | | | | X Consult with sponsor medical monitor | Yes |

AE, adverse event; CTCAE, Common Terminology Criteria for Adverse Events, version 4.03; HRV, Hypersensitivity Reaction Visit; NCI, National Cancer Institute.

<sup>&</sup>lt;sup>a</sup> NCI-CTCAE grade determination is performed by the investigator and may be done either via telephone or clinic visit.

<sup>&</sup>lt;sup>b</sup> The investigator will instruct the subject to maintain the rAvPAL-PEG dose at the time of AE onset until improvement to grade 1 or resolution (per investigator assessment in the clinic or via telephone).

<sup>&</sup>lt;sup>e</sup>The rAvPAL-PEG dose may be reduced or interrupted if necessary per investigator determination.

<sup>&</sup>lt;sup>d</sup> If a subject has an NCI-CTCAE grade ≥3 hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor, the subject may be permanently discontinued from study drug.

<sup>&</sup>lt;sup>c</sup> If the investigator determines that the NCI-CTCAE grade ≥3 hypersensitivity AE is related to administration with rAvPAL-PEG, the subject will be asked to return to the clinic within 24 hours of event onset for evaluation, including laboratory tests (chemistry, hematology, urinalysis, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE [sampling must be performed >8 hours after event onset and before the next dose of study drug], urine albumin/creatinine ratio, urinary N-methyl histamine, CRP, C3, C4, and tryptase).



# 9.1.1.3 Response to Anaphylaxis

If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and tryptase (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then be made whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose level.

For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equipment for emergency resuscitation (including epinephrine) within easy access. The subject must be observed for 30 minutes following administration due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and NSAIDs approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. NSAIDs should be given with food and may be omitted if not tolerated.

# 9.1.2 Study Stopping Criteria

If an NCI-CTCAE grade  $\geq$  3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening or required treatment to prevent a life-threatening event:

- Cyanosis or  $SpO_2 \le 92\%$
- Hypotension with SBP < 90 mm Hg (adults)
- Neurologic alteration: loss of consciousness, collapse, incontinence

Brown's severity criteria are presented in Table 9.1.2.1.



Table 9.1.2.1: Brown's Severity Criteria

| Brown's Criteria for | |
|---|---|
| Hypersensitivity Reactions | Definition |
| Mild (1) | Generalized erythema, urticaria, periorbital edema, or angioedema |
| skin and subcutaneous tissue | |
| Moderate (2) | Dyspnea, stridor, wheeze, nausea, vomiting, dizziness (pre-syncope), |
| features suggested respiratory, | diaphoresis, chest or throat tightness, or abdominal pain |
| cardiovascular, or | |
| gastrointestinal involvement | |
| Severe (3) | Cyanosis or SpO <sub>2</sub> ≤ 92% at any stage, hypotension (SBP < 90 mm Hg in |
| hypoxia or neurologic | adults), confusion, collapse, loss of consciousness, or incontinence |
| compromise | |

#### 9.1.3 **Dose Modifications**

## 9.1.3.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events for an individual subject. Dose increases >350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.




# 9.1.3.2 Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse event (any hypersensitivity reaction as defined in Section 9.1.1). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be adjusted.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L ), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

# 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

## 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.




- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use two acceptable methods of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

## 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the sponsor's medical monitor. However, subjects who discontinued from study drug early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).




- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG necessitating early termination from a previous rAvPAL-PEG study or known hypersensitivity to any of its excipients.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

## 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study drug should continue to perform the study tests and evaluations until study completion. For subjects who discontinue from the study, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study drug include, but are not limited to, the following:

- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy and refer to Section 9.1 for details on re-introduction of study drug following pregnancy and breastfeeding).

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.




If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

## 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in their previous rAvPAL-PEG study. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.

## 9.4 Treatments

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies will be dosed with the same or higher dose that was administered upon completion of that study provided that there was no interruption in dosing. rAvPAL-PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be adjusted per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects may be eligible to self-administer study drug if he or she meets the following criteria:




- The subject has no cognitive impairments that may increase the safety risk of self-administration per the assessment of the investigator.
- The subject has been approved for self-administration of study drug by the sponsor's medical monitor.
- The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely.
- The subject has been provided with two epinephrine injectors and has been trained on when and how to administer it. The subject will be instructed to carry one epinephrine injector with them at all times.

Qualified study site personnel will train each eligible subject on all procedures for self-administration of study drug (vial and syringe and prefilled syringe drug products) under the supervision of the PI. Qualified study site personnel will also be required to observe the subject prepare and perform at least 1 injection prior to allowing the subject to self-administer a dose at home. The subject will see a study site nurse or home healthcare nurse in person every week or receive a telephone call from site staff to ensure that the subject continues to perform all self-administration procedures correctly, to assess adverse events, and to answer questions throughout the duration of the study. The study site nurse or home healthcare nurse will also perform the regularly scheduled assessments and procedures as outlined in Table 9.1.1 and Section 12; the subject must perform a clinic visit monthly at minimum. Training materials and other information specific to the study site personnel are provided in the Subject Self-Administration Training Materials. Prefilled syringes are dispensed to subjects only after the subject (or caregiver) has completed training and competency is demonstrated in the clinic. Additional regular refresher training occurs in the clinic, every 24 weeks, and more often as needed.

Subjects who are eligible for self-administration will be provided with a Subject Study Manual. Self-administration training materials will be provided in the Subject Study Manual to supplement the in-person training provided by the qualified study site personnel. The Subject Study Manual will include step-by-step instruction on the following:

- How to prepare and perform the injections of study drug safely.
- How to receive, track, store, prepare, and return both used and unused study drug.
- How to safely use and dispose of syringes, including prefilled syringes, used for injections of study drug.
- How to use a new syringe and vial or new prefilled syringe every time drug is administered.



- How to care for their injection site after an injection of study drug.
- How to identify an adverse reaction and how to report this reaction to the study site.
- How and when to use epinephrine injectors.
- Who to contact at the study site in case of an emergency.

The PI or the sponsor's medical monitor may request that self-administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse.

Subjects who are within the target Phe range may also be permitted to convert from weight-based dosing to fixed dosing (refer to Section 9.4.4).

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site or subject with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplying the study drug to subjects who qualify for self-administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites.

Information regarding supplying study drug to subjects who qualify for self-administration is provided in the Subject Self-Administration Training Materials.

## 9.4.2 Identity of Investigational Product (IP)

## 9.4.2.1 Product Characteristics and Labeling

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self-administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5±0.2 mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

Or

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8±0.3 mL to deliver 20 mg of rAvPAL-PEG per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8±0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

|----------|------------|---------|
|----------|------------|---------|

Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Table 9.4.2.1.1: Prefilled Syringe Volume, Concentration, and Dose

| Prefilled Syringe | Volume | Concentration | Dose |
|-------------------|--------|---------------|--------|
| Sku #1 | 0.5 mL | 5 mg/mL | 2.5 mg |
| Sku #2 | 0.5 mL | 20 mg/mL | 10 mg |
| Sku #3 | 1.0 mL | 20 mg/mL | 20 mg |

Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be eligible to transition from vial and syringe to prefilled syringe dosing. Additionally, regular refresher training on use of prefilled syringe will be provided in study clinic every 24 weeks, and more often as needed.

Subjects should convert their vial and syringe dose to prefilled syringe dose using the following table:




Table 9.4.2.1.2: Conversion from Vial and Syringe Dose to Prefilled Syringe Dose

| Daily Dose (mg)<br>Range | Daily Dose (mg)<br>Round To <sup>a</sup> | # of 2.5mg<br>Prefilled Syringe<br>Needed | # of 10mg<br>Prefilled Syringe<br>Needed | # of 20mg<br>Prefilled Syringe<br>Needed |
|---|---|---|---|---|
| 0 - 3.7 | 2.5 | 1 | 0 | 0 |
| 3.8 - 6.2 | 5 | 2 | | |
| 6.3 - 8.7 | 7.5 | 3 | | |
| 8.8 – 11.2 | 10 | | 1 | |
| 11.3 - 13.7 | 12.5 | 1 | 1 | |
| 13.8 - 16.2 | 15 | 2 | 1 | |
| 16.3 – 18.7 | 17.5 | 3 | 1 | |
| 18.8 - 21.2 | 20 | | | 1 |
| 21.3 - 23.7 | 22.5 | 1 | | 1 |
| 23.8 - 26.2 | 25 | 2 | | 1 |
| 26.3 – 28.7 | 27.5 | 3 | | 1 |
| 28.8 – 31.2 | 30 | | 1 | 1 |
| 31.3 - 33.7 | 32.5 | 1 | 1 | 1 |
| 33.8 – 36.2 | 35 | 2 | 1 | 1 |
| 36.3 – 38.7 | 37.5 | 3 | 1 | 1 |
| 38.8 – 41.2 | 40 | | | 2 |
| 41.3 – 44.9 | 42.5 | 1 | | 2 |
| 45 – 54.9 | 50 | | 1 | 2 |
| 55 – 64.9 | 60 | | | 3 |
| 65 - 74.9 | 70 | | 1 | 3 |
| 75 – 84.9 | 80 | | | 4 |
| 85 – 94.9 | 90 | | 1 | 4 |
| 95 – 104.9 | 100 | | | 5 |
| 105 – 114.9 | 110 | | 1 | 5 |
| 115 – 124.9 | 120 | | | 6 |
| 125 – 134.9 | 130 | | 1 | 6 |
| 135 – 144.9 | 140 | | | 7 |
| 145 – 154.9 | 150 | | 1 | 7 |

<sup>&</sup>lt;sup>a</sup> For <45 mg/day, round to nearest 2.5 mg; for ≥45 mg/day, round to nearest 10 mg.


The excipients in this drug product wre tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60 600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity AE) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

For vial and syringe, drug product packaging will be identified with the lot number and expiration date and will be provided in a box labeled with the study number.

For prefilled syringe, drug product packaging will be identified with the size (2.5 mg, 10 mg, or 20 mg), lot number, and kit identification (ID). The expiration date will be available in a separate Certificate of Compliance issued for each lot.

# 9.4.3 Storage

IP must be stored at  $5 \pm 3$  °C ( $41 \pm 5$  °F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

Specific instructions for storage of study drug for subjects who qualify for self-administration are provided in the Subject Self-Administration Training Materials.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg (or 375 mg for subjects receiving a fixed dose).

For subjects receiving weight-based dosing, dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to



accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of  $60\text{-}600 \,\mu\text{mol/L}$  for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information presented in Table 9.4.4.1.

Table 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen

| Weight-based dose (mg/kg) | Equivalent fixed dose (mg) | Vol for 15 mg/ml concentration (ml) (vial) <sup>a</sup> |
|---|---|---|
| 0.03 | 2.5 | 0.17 |
| 0.06 | 5 | 0.33 |
| 0.12 | 10 | 0.67 |
| 0.25 | 20 | 1.33 |
| 0.5 | 40 | 2.67 |
| 1.0 | 75 | 5 |
| 2.0 | 150 | 10 |
| 3.0 | 225 | 15 |
| 4.0 | 300 | 20 |
| 5.0 | 375 | 25 |

<sup>&</sup>lt;sup>a</sup> Applies to both 1.0 and 1.3 ml withdrawal.

It is preferable that the injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff, other qualified and trained study personnel, or qualified subjects.




Information for dosing of subjects who enroll into this study after completing previous rAvPAL studies is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10.

Instructions for administration of study drug for subjects who qualify for self-administration are provided in the Subject Self-Administration Training Materials.

## 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in their previous rAvPAL-PEG study.

## 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study.

## 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered by clinic staff or other qualified and trained study personnel.

Subjects may self-administer study drug at home if approved by the sponsor's medical monitor and if adequate training is provided (refer to Section 9.4).

## 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the sponsor's medical monitor must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in a previous rAvPAL-PEG study) or investigational medical device within 30 days before Screening, or




requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior hypersensitivity AE to rAvPAL-PEG or a PEG-containing product will be encouraged to be premedicate as outlined in Section 9.1.1. If the hypersensitivity AE worsens with a repeat injection (as determined by the Investigator in consultation with the sponsor's medical monitor) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior hypersensitivity AE to rAvPAL-PEG or a PEG-containing product may participate in this study (refer to Section 9.3.2).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

# 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

### 9.4.10 Dose Interruption and Missed Doses

Information for dosing of subjects who enroll into this study after completing previous rAvPAL-PEG studies is provided in Section 9.1.

During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator. After a dosing interruption of ≥ four consecutive doses, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first week of dosing of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30 minutes following administration due to restarting dosing. Premedication with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs) approximately 2-3 hours prior to study drug should be administered following any dose interruption of ≥ four consecutive doses. NSAIDs should be given with food and may be omitted if not tolerated. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects



should continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 9.1.1) during any dosing interruption.

Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study drug per discretion of the Sponsor or Investigator (refer to Section 9.3.3).

# 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), IP returned, and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

## 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

Subjects who qualify for self-administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials).

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

## 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator.



A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next monthly study visit. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4.

## 9.7 Efficacy and Safety Variables

## 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

|----------|------------|---------|
|----------|------------|---------|

**Table 9.7.1.1: Summary of Laboratory Assessments** 

| Laboratory Assessment | Party Responsible for<br>Performing Test | Section in Protocol for Details |
|---|---|---|
| Clinical laboratory tests | Central laboratory | 9.7.6 |
| Antibody testing | BioMarin <sup>a</sup> or CRO | 9.7.5.2 |
| PK variables | BioMarin | 9.7.3 |
| Blood Phe concentrations | Central laboratory | 9.7.2.1 |
| Pregnancy test (urine) and sedimentation rate | Local laboratory | 9.7.6,<br>9.7.5.1 |
| Urinalysis | Central laboratory | 9.7.6 |

Phe, phenylalanine; PK, pharmacokinetic.

## 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, including allergy history, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

## 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.

### 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. Weight will be measured at Screening and then monthly.

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL IgE and anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



### 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the Final Follow-Up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

### **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Screening, Week 48, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

## 9.7.2 Efficacy Variable

## 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn monthly, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1).

Blood Phe may be collected more often than monthly at the discretion of the Investigator should more frequent monitoring of blood Phe levels be clinically required.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Subjects enrolled in the Substudy will have additional PK sampling performed. For subjects participating in the Substudy, PK sampling will be performed as follows:

- For subjects who are administered rAvPAL-PEG once per week, plasma PK sampling will be performed pre-dose and every 24 hours thereafter (24, 48, 72, and 96 hours if possible), and then pre-dose of the next weekly dose.
- For subjects who are administered rAvPAL-PEG two or three times per week, plasma PK sampling will be performed pre-dose and every 24 hours during the longest period between doses, when possible, and then pre-dose of the next dose.
- For subjects who are administered rAvPAL-PEG four to seven times per week, plasma PK sampling will be performed pre-dose and every 12 hours during the longest period between doses, when possible, and then pre-dose of the next dose.

See Table 9.1.2 for additional details.

BioMarin will perform the analysis.



## 9.7.4 Exploratory Efficacy Variable

Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits on a monthly basis. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each month. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator.

### 9.7.5 Safety Variables

## 9.7.5.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 9.1.1). Female subjects with a positive serum pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

## 9.7.5.2 Antibody Testing

Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1). Immunogenicity assays will be performed at the time points indicated in the Schedule of Events (Table 9.1.1).

BioMarin or CRO will perform all anti-body testing, except for IgE antibodies, which will be assessed by a Contract Research Organization.

## 9.7.6 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant.



All abnormal clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the abnormal result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.




# **Table 9.7.6.1: Clinical Laboratory Tests**

| Blood Chemistry | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if |
| Alkaline Phosphatase | Hematocrit | Color | - applicable <sup>a</sup> |
| ALT (SGPT) | WBC count | рН | Phenylalanine |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Sedimentation rate <sup>a</sup> |
| BUN | Differential cell count | Protein | |
| Creatinine | | Glucose | |
| GGT | | Spot urine albumin/creatinine ratio | Additional Unscheduled<br>Hypersensitivity Reaction<br>Visit Tests <sup>b</sup> |
| Total protein | | Nitrite | CH50 |
| Calcium | | Urobilinogen | $C_1, C_3, C_4$ |
| Sodium | | Hemoglobin | Serum tryptase level <sup>b</sup> |
| Potassium | | Bilirubin | CRP |
| Glucose | | | Urine N-methyl histamine |
| | | | Urine albumin/creatinine ratio |
| Uric acid | | | Complement Testing <sup>c</sup> |
| CO <sub>2</sub> | | | C <sub>3</sub> |
| Chloride | | | C <sub>4</sub> |

ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; C, complement; CH50, total hemolytic complement; CO2, carbon dioxide; CRP, C-reactive protein; GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.

<sup>&</sup>lt;sup>a</sup> To be performed by central laboratory. If urine pregnancy test is positive or equivocal, serum sample will be taken and assessed by a central laboratory.

<sup>&</sup>lt;sup>b</sup> Perform within 24 hours of event onset.

<sup>&</sup>lt;sup>c</sup> Complement C<sub>3</sub> and C<sub>4</sub> to be drawn at the Screening Visit and then quarterly or as needed to resolve abnormal test results.



#### 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a subject administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment run-in).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The study AE reporting period is as follows: After informed consent but prior to initiation of study drug, only SAEs associated with any protocol-imposed interventions will be reported. After informed consent is obtained and the first administration of study drug, all non-serious AEs and SAEs reporting period begins and continues until 4 weeks following the last administration of study drug or the Study Completion Visit/Early Termination Visit, whichever occurs last (refer to Section 12). The criteria for determining, and the reporting of SAEs is provided in Section 10.2.

For this study, a medical device is defined as the prefilled syringe and all of the component parts. The reporting period for device-related events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe. Events assessed by the investigator as related to the device, including malfunction, injury, or medication error, will be captured into an electronic data capture system. All serious events related to the device will be reported to BioMarin Pharmacovigilance (BPV) within 24 hours using the device-related event report form and entered onto the appropriate eCRF page(s) as required.



The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study drug or study participation is not the cause of the AE. Outcome of AEs (and resolution dates) should be documented on the appropriate CRF page(s) and in the subject's medical record unless the subject is lost to follow-up or it has been determined that the study drug or study participation is not the cause of the AE.

The Investigator responsible for the care of the subject or qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to seriousness, which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the severity of each AE using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.

| Grade | Description |
|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life-threatening: hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL) <sup>b</sup> |
| 4 | Life threatening or debilitating: consequences; urgent intervention indicated |
| 5 | Death related to AE |

Grade 4 and 5 AEs should always be reported as SAEs.

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

<sup>&</sup>lt;sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.



The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR |
| | The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly<br>Related | The administration of the IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably | The administration of IP and the occurrence of the AE are reasonably related in time |
| Related | AND |
| | The AE is more likely explained by exposure to the IP than by other factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).

#### **10.2** Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Is fatal.
- Is life threatening.
  - Note: Life-threatening refers to an event that places the subject at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires or prolongs inpatient hospitalization.
- Results in persistent or significant disability or incapacity.
- Is a congenital anomaly or birth defect in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.




 Important medical events or reactions that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes above should also usually be considered serious.

For this protocol, anaphylaxis per NIAID/FAAN criteria for the clinical diagnosis of anaphylaxis is designated as an AE of special interest (serious or nonserious and irrespective of severity) to facilitate rapid reporting and sponsor review. All occurrences of anaphylaxis per NIAID/FAAN criteria will be reported to the sponsor within 24 hours of the site becoming aware of the event using the SAE form. Severity and serious criteria (if applicable) should be reported on the SAE form.

The reporting period for SAEs related to protocol imposed interventions begins after informed consent is obtained, the reporting period for all SAEs begins after first dose of study drug and continues until 4 weeks following the last administration of study drug or End of Treatment Visit. The reporting period for Serious Device Related Events begins after first dose of study drug and ends with the last administered dose.

All SAEs (including serious device-related events), whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form or device Report Form to BioMarin Pharmacovigilance (BPV). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study drug or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the subject's medical record.

For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).

At the last scheduled visit, the Investigator should instruct each subject to report any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study drug.

The Investigator should notify the study Sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior

Amendment 7: 16 December 2015




study drug. The Sponsor should also be notified if the Investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that participated in this study.

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

# 10.3 Pregnancy

Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. The reporting period for pregnancies begins with informed consent and continues until 4 weeks following the last study drug dose. In addition, pregnancy in a subject is also reported on the End of Study CRF if the subject withdraws from the study due to pregnancy. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution to BPV in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

### **10.4** Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "... in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours.



Examples of situations that may require urgent safety measures include discovery of the following:

- Immediate need to revise the IP administration (i.e., modified dose amount or frequency not defined in protocol).
- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.

## 10.5 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the Sponsor's Medical Office sponsor's medical monitor r any AEs for which the issue of seriousness is unclear or questioned. Contact information for the sponsor's medical monitor is as follows:

Name: , MD Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:

Fax:

E-mail:



#### 11 APPROPRIATENESS OF MEASUREMENTS

## 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

## 11.2 Diet Diary

A 3-day diet diary will be issued to subjects for completion and will be brought to clinic on a monthly basis for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6.



#### 12 STUDY PROCEDURES

### 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

## 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Chest X-ray
- 12-lead ECG
- Clinical laboratory tests (including spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis)
- Complement C<sub>3</sub> and C<sub>4</sub>
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in a previous rAvPAL-PEG study, these assessments may be the same as those used for the last visit of the previous study, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications




assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. If there is a skin reaction that lasts  $\geq$  14 days, the Skin Reaction eCRF should be completed. A photograph of the skin reaction may be taken by the subject or the site to help assess the event and may be collected by the sponsor.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done daily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

## 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator)

#### 12.3.2 Weekly Telephone Visit

Subjects should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit:

- Injection-site self inspection (previous and current injection site)
- Assessment of AEs



- Concomitant medications
- Confirmation of dose level, frequency, and study drug administration

## 12.3.3 Substudy Visits

For subjects participating in the PK substudy, refer to Section 9.7.3 and Table 9.1.2.

# 12.3.4 Monthly Visits (Week 4, 8, 12, etc)

Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Beginning with Week 4, monthly visits must be performed in the clinic. The following study activities will be performed:

- Vital signs
- Weight
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) For safety reasons, this test must be performed prior to the chest X-ray.
- Chest x-ray (Week 48 visit only)
- Assessment of AEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.)
- Prefilled syringe self-administration training (to be performed prior to subjects transitioning from vial and syringe drug product to prefilled syringe drug product).
- Administer study drug
- If additional training is needed on days subsequent to the monthly visit, additional clinic visit(s) or HHRN may be used.

Amendment 7: 16 December 2015

# 12.3.5 Quarterly Visits (Week 12, 24, 36, etc)

Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.




Beginning with Week 12, quarterly visits consist of all monthly (Section 12.3.4) activities listed above as well as the additional study activities listed below:

- Physical examination
- Complement C<sub>3</sub> and C<sub>4</sub>
- Sedimentation rate
- PK sample
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Prefilled syringe refresher training (every 24 weeks only)

# 12.3.6 Unscheduled Hypersensitivity Reaction Visit

Subjects who have an NCI-CTCAE grade  $\geq 3$  hypersensitivity reaction after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 24 hours) the reaction.

- Vital signs
- Clinical laboratory tests
- Urine/albumin creatinine ratio
- CRP, CH50, C1, C3, and C4
- Urine N-methyl histamine
- Serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only (performed > 8 hours after event onset)
- Serum tryptase level
- Skin biopsy (optional; affected and not affected area; to be performed within 1 week of the reaction)
- Assessment of AEs
- Concomitant medications

Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects may resume study drug administration per the discretion of the Principal Investigator and the sponsor's medical monitor.

### 12.4 Study Completion/Early Termination Visit

Subjects should perform the Study Completion Visit 4 weeks after the last dose of study drug




or after completion of study participation, whichever occurs last.

For subjects who terminate from the study early (refer to Section 9.3.3), the Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug or after withdrawal from study participation, whichever occurs last. Subjects who terminate from study drug early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)



## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

### 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

## 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF).

The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics of vital signs, physical examination results, ECG results, and X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

#### 14.3 Pharmacokinetic Analysis

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $C_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F). Should



data become available from previous rAvPAL-PEG studies that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

### 14.3.1 Pharmacokinetic Substudy Analysis

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored. This substudy has been completed as of 20 December 2013.

## 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the SAP) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis.

Details regarding exploratory analyses will be provided in the Statistical Analysis Plan.

#### 14.5 Determination of Sample Size

Subjects who participated in previous rAvPAL-PEG studies may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

#### 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.



### 14.7 Interim Analyses

Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

## 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.



### 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Assess the effect and relevance of new external evidence.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.2.
- Make recommendations to the BioMarin concerning continuation or termination of the study or other study modifications based on observations.



### 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment, unless the executed Clinical Trial Agreement between BioMarin and the institution of the investigator specifies otherwise. If the subject has followed the Investigator's instructions, BioMarin may pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.



#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. Upon completion of the clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.



#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (e.g., subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.



#### 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages the publication of these data in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Trial Agreement between BioMarin and the Investigator/Institution. Consideration for authorship of all publications will be based on compliance with the Uniform Requirements for Manuscripts Submitted to Biomedical Journals ("Uniform Requirements") of the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org/about-icmje/faqs/icmje-recommendations/) and good publication practices (GPP).



#### 21 REFERENCES

Armstrong, JK, Hempel, G, Koling, S, Chan, LS et. al. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007

Brown, SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 114[2], 371-376. 2004

Chen, AM, Scott, MD. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001

Davis, S, Abuchowski, A, Park, YK, Davis, FF. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981

Fisch, RO. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000

Gamez, A, Wang, L, Sarkissian, CN, Wendt, D et. al. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007

Ganson, NJ, Kelly, SJ, Scarlett, E, Sundy, JS et. al. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006

Guttler, F, Azen, C, Guldberg, P, Romstad, A et. al. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003

Harris, JM, Chess, RB. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003

Huttenlocher, PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000

Judge, A, McClintock, K, Phelps, JR, Maclachlan, I. Hypersensitivity and loss of disease site targeting caused by antibody responses to PEGylated liposomes. Mol Ther 13[2], 328-337. 2006

Kaufman, S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989

Koch, R, Hanley, W, Levy, H, Matalon, K et. al. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003




Lapis. Long-term Correction of PKU in the Pahenu2 Mouse by Mutant and Chemically Modified Forms of Phenylalanine Ammonium Lyase. ASHG 57th Annual Meeting The American Society of Human Genetics) 2007.

Lee, PJ, Lilburn, M, Baudin, J. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003

Levy, HL. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003

Matalon, R, Surendran, S, Matalon, KM, Tyring, S et. al. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003

Richter, AW, Akerblom, E. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983

Richter, AW, Akerblom, E. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984

Rouse, B, Azen, C. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004

Sampson, HA, Munoz-Furlong, A, Campbell, RL, Adkinson, NF, Jr. et. al. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol 117[2], 391-397. 2006

Scott, MD, Murad, KL, Koumpouras, F, Talbot, M et. al. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997

Scriver, CR, Kaufman. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-1724.

Walter, JH, White, FJ, Hall, SK, MacDonald, A et. al. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002

Webster, R, Didier, E, Harris, P, Siegel, N et. al. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007



#### 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.


# 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003, Amendment 7

| Investigator Signature | Date |
|------------------------|------|
| Printed name: | |

# Accepted for the Sponsor:

| | 1(0 | DEC 2015 |
|---------------------------|-----|----------|
| Medical Monitor Signature | | Date |
| Printed name: | | |

|----------|------------|---------|
|----------|------------|---------|

#### 24 PROTOCOL AMENDMENT TEXT REVISIONS

The following is a summary of significant protocol revisions; added text is <u>underlined</u> and deleted text is <u>struck</u>. The study design schematic (Figure 9.1.1) and Schedule of Events (Table 9.1.1) were revised accordingly. Additional administrative changes have been made for consistency and clarity throughout this amendment and are reflected in the protocol body. Revisions made to the Synopsis (Section 2) are reflected in the corresponding protocol section as appropriate. Revisions to cross references to protocol tables, figures, sections, and references reside within the protocol body.

| Section | Davision | Rationale for |
|---|---|---|
| Section Section 2, Section 9.1, Study Design | Because the risks of taking rAvPAL-PEG during pregnancy and breastfeeding are unknown, subjects cannot take rAvPAL-PEG if they are trying to conceive, are pregnant, or are breastfeeding. Male subjects who are planning to impregnate a female partner and female subjects who are trying to become pregnant during the study will be discontinued immediately from study drug. Male subjects who have impregnated a female partner may re-start study drug after conception but must return to the study-required contraception use, which must include one barrier method. Subjects who remain in the study after discontinuation of study drug due to pregnancy may re-introduce rAvPAL-PEG dosing after the birth has been reported (or termination of the pregnancy) and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to conceive. Re-starting rAvPAL-PEG dosing must be per investigator and sponsor agreement based on an assessment of the known risks and potential benefits while taking BMN 165. Female subjects must return to the study-required contraception use, which must include one barrier method, immediately after the birth (or termination of the pregnancy). | Change 2 |
| Section 2, Section 9.3.1,<br>Inclusion Criteria | Individuals eligible to participate in this study must meet all of the following criteria: • Sexually active subjects must be willing to use <a href="mailto:antwo">antwo</a> acceptable methods of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study. | 3 |
| Section 2, Duration of Treatment | Up to <u>102</u> 98 months. | 4 |
| Section 9.1, Study Design | Because the risks of taking rAvPAL-PEG during pregnancy and breastfeeding are unknown, subjects cannot take rAvPAL-PEG if they are trying to conceive, are pregnant, or are breastfeeding (refer to Section 9.3.2, Exclusion Criteria). Male subjects who are planning to impregnate a female | 2 |

|----------|------------|---------|
|----------|------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | partner and female subjects who are trying to become pregnant during the study will be discontinued immediately from study drug. Male subjects who have impregnated a female partner may re-start study drug after conception but must return to the study-required contraception use (refer to Section 9.3.1, Inclusion Criteria), which must include one barrier method. Subjects who remain in the study after discontinuation of study drug due to pregnancy may re-introduce rAvPAL-PEG dosing after the birth has been reported (or termination of the pregnancy) and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to conceive. Re-starting rAvPAL-PEG dosing must be per investigator and sponsor agreement based on an assessment of the known risks and potential benefits while taking BMN 165. Female subjects must return to the study-required contraception use (refer to Section 9.3.1), which must include one barrier method, immediately after the birth (or termination of the pregnancy). | |
| Table 9.1.1, Schedule of Events | The table has been updated to reflect changes made with this amendment. | 1, 5, 6 |
| Section 9.3.3, Removal of<br>Subjects from Treatment<br>or Assessment | Reasons for which the Investigator or BioMarin may withdraw a subject from the study treatment drug include, but are not limited to, the following: • Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy and refer to Section 9.1 for details on re-introduction of study drug following pregnancy and breastfeeding). | 2 |
| Section 10.1, Adverse<br>Events | After informed consent is obtained and the first administration of study drug, all non-serious AEs and SAEs reporting period begins and continues until 4 weeks following the last administration of study drug or the Study Completion Visit/Early Termination Visit, whichever is longeroccurs last (refer to Section 12). The criteria for determining, and the reporting of SAEs is provided in Section 10.2. | 5 |
| Section 10.3, Pregnancy | Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. The reporting period for pregnancies begins with informed consent and | 2 |

|----------|------------|---------|
|----------|------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | continues until 4 weeks following the last study drug dose. In addition, pregnancy in a subject is | |
| | also reported on the End of Study CRF if the subject withdraws from the study due to pregnancy | |
| Section 12.3, Treatment<br>Period | During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. All study activities will occur on the first day of each week unless otherwise noted. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. If there is a | 1 |
| | skin reaction that lasts ≥14 days, the Skin Reaction eCRF should be completed. A photograph of the skin reaction may be taken by the subject or the site to help assess the event and may be collected by the sponsor. | |
| Section 12.4, Study<br>Completion/Early<br>Termination Visit | Subjects should perform the Study Completion Visit 4 weeks after the last dose of study drug or after completion of study participation, whichever occurs last. For subjects who terminate from the study early (refer to Section 9.3.3), tThe Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug or after withdrawal from study participation, whichever occurs last | 5 |
| Section 20, Use of<br>Information and<br>Publication | BioMarin recognizes the importance of communicating medical study data and therefore encourages the publication of these data in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Trial Agreement between BioMarin and the Investigator/Institution. Consideration for authorship of all publications will be based on compliance with the Uniform Requirements for Manuscripts Submitted to Biomedical Journals ("Uniform Requirements") of the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org/about-icmje/faqs/icmje-recommendations/) and good | 6 |

|----------|------------|---------|
|----------|------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | publication practices (GPP). | |
| | BioMarin recognizes the importance of communicating medical study data and therefore | |
| | encourages their publication in reputable scientific journals and at seminars or conferences. The | |
| | details of the processes of producing and reviewing reports, manuscripts, and presentations based | |
| | on the data from this study will be described in the Clinical Trial Agreement between BioMarin and | |
| | the institution of the investigator. | |



### **CLINICAL STUDY PROTOCOL**

Study Title: Long-term Extension of a Phase 2, Open-Label, Dose-Finding

Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with

**PKU** 

Protocol Number: PAL-003

Investigational Product: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis

phenylalanine ammonia lyase)

IND/EUDRACT Number: IND 076269

Indication: Phenylketonuria (PKU)

Sponsor: BioMarin Pharmaceutical Inc.

105 Digital Drive Novato, CA 94949

Development Phase: Phase 2

Sponsor's Responsible Medical

Monitor:

MS

Duration: Approximately 119 months

Dose: 0.001 to a maximum weekly dose of 5.0 mg/kg or 375 mg/week

Date of Original Protocol:

October 08, 2008

Date of Amendment 1:

February 09, 2009

Date of Amendment 2:

October 30, 2009

Date of Amendment 3:

May 04, 2011

Date of Amendment 4:

June 7, 2012

Date of Amendment 5: February 28, 2014
Date of Amendment 6: October 30, 2014
Date of Amendment 7: December 16, 2015

Date of Amendment 8: March 31, 2017


May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin. This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.

BioMarin is a registered trademark of BioMarin Pharmaceutical Inc.




#### CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Amendment: 8

**Date: 31 March 2017** 

#### RATIONALE AND SUMMARY OF CHANGES

This section provides a numbered list of all significant changes and supporting rationale:

- 1. To monitor subject safety, a repeat urinalysis should be performed for subjects who have an abnormal or elevated proteinuria test result. Additionally, first or second morning void is being recommended for all urinalyses collected during the study. In addition, information regarding renal toxicity due to exposure to PEG has been updated in the background section (Section 7.4.1).
- 2. Additional instruction has been added for subjects who are pregnant or are planning to become pregnant (or impregnate a female partner) during the study for clarity and to monitor subject safety.
  - Subjects who are planning to conceive must stop study drug at least
     4 weeks prior to trying to conceive and must use two forms of acceptable contraception prior to trying to conceive.
  - Subjects who are planning to become pregnant (or impregnate a female partner) during the study may modify their diet in consultation with the investigator and/or study dietician.
  - Subjects who are pregnant or are trying to conceive and have temporarily discontinued study drug are not required to perform the scheduled pharmacokinetic (PK) assessments.
  - O Subjects who have been confirmed to be pregnant with a serum pregnancy test are not required to perform the urine pregnancy tests while pregnant.
  - Upon re-starting study drug following a pregnancy or breastfeeding, female subjects must have a confirmed negative urine pregnancy test result.
- 3. Additional instruction regarding adverse event (AE) and serious AE (SAE) reporting has been added to provide clarity and to improve the quality of safety reporting. The following have been added:
  - Guidance on factors suggestive of a causal relationship to study drug to facilitate investigator assessments of AEs
  - o Guidance on how to report AEs occurring secondary to other events
  - o Guidance on reporting of persistent versus recurrent AEs




- Guidance on when abnormal laboratory test results should be reported as AEs
- O Guidance on how pre-existing conditions should be recorded
- Guidance on where and how physician examination findings should be reported as AEs
- Guidance on scenarios that do not require reporting hospitalization as an SAE
- Guidance on how to report deaths
- Guidance on how to report abortions
- o Guidance on reporting post-study SAEs
- O Guidance regarding sponsor request for additional case details for SAEs and AEs of special interest, including hospital discharge, consultant reports, and autopsy reports
- 4. To monitor for subject safety, subjects who have an elevated urine/albumin creatinine ratio (defined as confirmed result of ≥ 100 mg/g for subjects with results within normal range at baseline or a confirmed increase of 100-200 mg/g from baseline for subjects with elevated results at baseline) should be referred to a nephrologist for consultation.
- 5. To monitor for subject safety, subjects who experience an injection-site skin reaction that lasts ≥14 days should be referred for a dermatology consultation and may be asked to perform a skin biopsy.
- 6. Instruction regarding the premedications to administer prior to injection of study drug has been revised to provide alternative medications to subjects who may not tolerate non-steroidal anti-inflammatory drugs (NSAIDS); subjects may alternatively be premedicated with antipyretics (eg, acetaminophen).
- 7. Information regarding exploratory sample analysis (use of leftover blood and urine samples) during the study and after the subject completes the study has been added.
- 8. The Schedule of Events has been modified; scheduled visits are to occur every 8 weeks (rather than every 4 weeks and quarterly) to align with the visit schedule in the ongoing extension (Part 4) of the Phase 3 study, 165-302.
- 9. The study duration has been extended from 102 months to approximately 119 months.
- 10. The responsible Medical Monitor has been changed.
- 11. Minor changes were made to improve clarity and consistency and update protocol language to reflect more recent information and/or instruction regarding study conduct.

| <b>B</b> OMARIN | PAL-003 A8 | Page 4 |
|-----------------|------------|--------|
|-----------------|------------|--------|

In addition, the Schedule of Events (Section 9.1) and Section 12 have been updated to reflect the changes in this amendment. Refer to Section 24 for a summary of the amendment revisions.



#### 2 SYNOPSIS

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| rAvPAL-PEG (PEGylated recombinant<br>Anabaena variabilis phenylalanine ammonia<br>lyase) | Reference: | |
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### TITLE OF STUDY:

Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU


**STUDY SITES**: Approximately 20 centers in the United States

**PHASE OF DEVELOPMENT**: Phase 2

#### STUDY RATIONALE:

The need exists for a treatment that will help individuals with phenylketonuria (PKU) safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits. This study is an extension of the rAvPAL-PEG Phase 2 studies PAL-002, PAL-004, and 165-205. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data were collected for subjects who have already achieved Phe reduction to within the protocol-defined target range. This substudy has been completed as of 20 December 2013.

|----------|------------|--------|
|----------|------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

## **OBJECTIVES**:

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objectives are as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.

### STUDY DESIGN AND PLAN:

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity is observed in a previous rAvPAL-PEG study. Subjects' doses will not exceed 375 mg/week.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the sponsor's medical monitor. The first dose will be administered in the clinic, and the subject must be observed for 30 minutes following administration. Additionally, subjects will be given two epinephrine injectors and will be instructed to carry one epinephrine injector with them at all times. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

| <b>BIOMARIN</b> | PAL-003 A8 | Page 7 |
|-----------------|------------|--------|
|-----------------|------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be reviewed with the clinical study staff on a monthly basis.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self-administration. Additional training will be provided to subjects and demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.

In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600  $\mu$ mol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points. After the subject's blood Phe concentration has been controlled to within a target range (60-600 µmol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator or Sponsor.
- The subject has completed the study through the Week 476 visit.
- The study is terminated.
- The study drug receives marketing authorization.

| <b>B</b> OMARIN | PAL-003 A8 | Page 8 |
|-----------------|------------|--------|
|-----------------|------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

Because the risks of taking BMN 165 during pregnancy and breastfeeding are unknown, subjects cannot take BMN 165 if they are trying to conceive, are pregnant, or are breastfeeding (refer to Section 9.3.2 for Exclusion Criteria). Male subjects who are planning to impregnate a female partner and female subjects who are trying to become pregnant during the study must be temporarily discontinued from study drug for 4 weeks prior to trying to conceive. During that time, subjects must use two acceptable methods of contraception. Subjects who are planning to become pregnant (or impregnate a female partner) may modify their diet in consultation with the investigator and/or study dietician. Subjects who are confirmed to be pregnant per a serum pregnancy test and are temporarily off study drug are not required to perform the scheduled urine pregnancy tests. Subjects who are pregnant or are trying to conceive and have temporarily discontinued study drug should not perform the scheduled PK assessments. Male subjects who have impregnated a female partner may re-start study drug after conception following the investigator's consultation with and approval by the medical monitor. Male subjects must return to the study-required contraception use, which must include one barrier method, prior to restarting study drug. Female subjects who remain in the study after temporary discontinuation of study drug due to pregnancy may restart BMN 165 dosing after a confirmed negative urine pregnancy test result, the birth has been reported (or termination of the pregnancy), and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to conceive. Re-starting BMN 165 dosing requires the investigator's prior consultation with and approval by the medical monitor. Female subjects must return to the study-required contraception use, which must include one barrier method, immediately after the birth (or termination of the pregnancy). Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not

#### PAL -003 Substudy

compromise subject safety.

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed. This substudy has been completed as of 20 December 2013.

| <b>B</b> OMARIN | PAL-003 A8 | Page 9 |
|-----------------|------------|--------|
|-----------------|------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| Anabaena variabilis phenylalanine ammonia lyase) NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### **Dose Modifications:**

### Dose Increase Methodology:

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations. An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4,0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events (any hypersensitivity reaction) for an individual subject. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.

#### Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower dose.

| <b>B</b> OMARIN | PAL-003 A8 | Page 10 |
|-----------------|------------|---------|
|-----------------|------------|---------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | 50.40.20.20.10.00.06.04 | |

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be adjusted.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30 µmol/L), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

#### **Safety Assessment Criteria:**

### **Response to Hypersensitivity Adverse Events**

Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. If non-steroidal anti-inflammatory medication (NSAIDs) is administered as a premedication, it should be given with food.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality. Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

### **Individual Stopping Criteria**

Subjects who have an NCI CTCAE grade  $\geq 3$  hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.




#### **Dosing in Response to Hypersensitivity Adverse Events**

Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG.

Once an AE (other than anaphylaxis) improves to grade 1 or resolves, study drug dose may be increased, maintained, or reduced. If dosing has been interrupted due to an AE (other than anaphylaxis) and the investigator determines it is safe for the subject to resume dosing, the first dose after improvement of the AE should be performed in the clinic. The subject must be observed for 30 minutes following administration due to restarting dosing. The subject may be advised to premedicate with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. If NSAIDs are administered as a premedication, they should be given with food.

# Response to Anaphylaxis

If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and tryptase (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then be made whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose level.

For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equipment for emergency resuscitation (including epinephrine) within easy access. The subject must be observed for 30 minutes following administration due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. If NSAIDs are administered as a premedication, they should be given with food.

## **Stopping Criteria:**

If an NCI-CTCAE grade ≥3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening or required treatment to prevent a life-threatening event:

- Cyanosis or  $SpO_2 \le 92\%$
- Hypotension with SBP < 90 mm Hg (adults)
- Neurologic alteration: loss of consciousness, collapse, incontinence

#### NUMBER OF SUBJECTS PLANNED:

Up to 100 subjects.

#### DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

Individuals eligible to participate in this study must meet all of the following criteria:

- Must have completed participation in a previous rAvPAL-PEG study.
- Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a

| <b>B</b> OMARIN | PAL-003 A8 | Page 12 |
|-----------------|------------|---------|
|-----------------|------------|---------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.

- Willing and able to comply with all study procedures.
- Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- Sexually active subjects must be willing to use two acceptable methods of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
- Maintained a stable diet.
- In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the sponsor's medical monitor. However, subjects who discontinued from study drug early due to a reaction are not eligible to enroll into this study.

| <b>B</b> OMARIN | PAL-003 A8 | Page 13 |
|-----------------|------------|---------|
|-----------------|------------|---------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

- Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- Concurrent disease or condition that would interfere with study participation or safety
  (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal,
  hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic,
  or psychiatric disease).
- Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- Known hypersensitivity to rAvPAL-PEG necessitating early termination from a previous rAvPAL-PEG study or known hypersensitivity to any of its excipients.
- Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- Creatinine > 1.5 times the upper limit of normal.

#### INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self-administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5 ± 0.2 mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

#### Or:

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8 ±0.3 mL to deliver 20 mg of rAvPAL-PEG per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8 ± 0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

| <b>B</b> OMARIN | PAL-003 A8 | Page 14 |
|-----------------|------------|---------|
|-----------------|------------|---------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

Or:

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be eligible to transition from vial and syringe to prefilled syringe dosing. Additionally, regular refresher training on use of prefilled syringe will be provided in study clinic every 24 weeks, and more often as needed.

The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL-PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu mol/L$ ), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu mol/L$  for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

#### **Fixed Dosing**

Subjects who have demonstrated efficacy (ie, blood Phe within the target range of 60-600 µmol/L for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week).

#### **DURATION OF TREATMENT:**

Approximately 119 months

# REFERENCE THERAPY(IES), DOSE, ROUTE AND REGIMEN:

None

#### **CRITERIA FOR EVALUATION:**

#### **Efficacy**:

Blood Phe concentrations will be measured.

### Immunogenicity:

| <b>B</b> OMARIN | PAL-003 A8 | Page 15 |
|-----------------|------------|---------|
|-----------------|------------|---------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase) | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | d' PEG L G |

The presence of antibodies (anti-PAL immunoglobulin G [IgG], anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-PEG neutralizing antibodies, anti-rAvPAL IgE, and anti-PEG-PAL IgE) will be assessed.

#### Safety:

Safety will be evaluated on the incidence of adverse events (AEs) and clinically significant changes in vital signs, ECG results, X-ray results, and laboratory test results.

#### Pharmacokinetic:

Plasma concentrations of rAvPAL-PEG will be measured for subjects participating in the Substudy.

#### **STATISTICAL METHODS:**

#### Sample Size:

Subjects who participated in a previous rAvPAL-PEG study may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

## **Safety Analysis**:

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by-subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics for vital signs, physical examination results, ECG results, X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

| <b>B</b> IOMARIN | PAL-003 A8 | Page 16 |
|------------------|------------|---------|
|------------------|------------|---------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 NAME OF FINISHED PRODUCT: rAvPAL-PEG (PEGylated recombinant Anabaena variabilis phenylalanine ammonia | SUMMARY TABLE Referring to Part of the Dossier: Volume: Page: Reference: | FOR NATIONAL<br>AUTHORITY USE<br>ONLY: |
|---|---|---|
| lyase) NAME OF ACTIVE INGREDIENT: phenylalanine ammonia lyase | | |

#### **Efficacy Analysis:**

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, standard deviation, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the Statistical Analysis Plan [SAP]) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

#### **Exploratory Analysis:**

Details regarding exploratory analyses will be provided in the SAP.

# **Substudy Analysis:**

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored.

#### **Pharmacokinetic Analysis:**

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $T_{max}$ ), half life ( $T_{max}$ ), and clearance ( $T_{max}$ ).




# 3 TABLE OF CONTENTS

| 1 | TIT | LE PAG | E | 1 |
|---|---|---|---|---|
| 2 | SYNOPSIS | | | |
| 3 | TABLE OF CONTENTS | | | |
| 4 | LIST | Γ OF AE | BBREVIATIONS AND DEFINITIONS OF TERMS | 21 |
| 5 | ETE | IICS | | 24 |
| | 5.1 | Institut | tional Review Board or Ethics Committee | 24 |
| | 5.2 | Ethical | Conduct of Study | 24 |
| | 5.3 | Subject | t Information and Informed Consent | 25 |
| 6 | INV | ESTIGA | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | 26 |
| 7 | INT | RODUC | CTION | 27 |
| | 7.1 | Noncli | nical Studies | 27 |
| | 7.2 | Previou | us Clinical Studies | 28 |
| | | 7.2.1 | Phase 1 Study, PAL-001 | 29 |
| | | 7.2.2 | Phase 2 Studies PAL-002, PAL-004, and 165-205 | 29 |
| | 7.3 | Study I | Rationale | 33 |
| | 7.4 | Summa | ary of Overall Risks and Benefits | 34 |
| | | 7.4.1 | Toxicity Due to Exposure to Polyethylene Glycol (PEG) | 34 |
| | | 7.4.2 | Immunologic Response | 35 |
| | | 7.4.3 | Management of Hypersensitivity Reactions | 37 |
| 8 | STU | DY OB | JECTIVES | 39 |
| 9 | INV | ESTIGA | ATIONAL PLAN | 40 |
| | 9.1 | Overal | l Study Design and Plan | 40 |
| | | 9.1.1 | Response to Hypersensitivity Adverse Events | 47 |
| | | 9.1.2 | Study Stopping Criteria | 49 |
| | | 9.1.3 | Dose Modifications | 50 |
| | 9.2 | Discus | sion of Study Design, Including Choice of Control Group | 51 |
| | 9.3 | Selecti | on of Study Population | 51 |
| | | 9.3.1 | Inclusion Criteria | 51 |
| | | 9.3.2 | Exclusion Criteria | 52 |

| BIO | MA | RIN | PAL-003 A8 | Page 18 |
|---|---|---|---|---|
| | 9.3.3 | Removal o | f Subjects from Treatment or Assessment. | 53 |
| | 9.3.4 | | entification and Replacement of Subjects | |
| | 9.4.1 | | Administered | |
| | 9.4.2 | | Investigational Product (IP) | |
| | 9.4.3 | | | |
| | 9.4.4 | | for Administration | |
| | 9.4.5 | Method of | Assigning Subjects to Treatment Groups | 61 |
| | 9.4.6 | | f Doses Used in the Study | |
| | 9.4.7 | | | |
| | 9.4.8 | Prior and C | Concomitant Medications | 61 |
| | 9.4.9 | Treatment | Compliance | 62 |
| | 9.4.10 | Dose Intern | ruption and Missed Doses | 62 |
| 9.5 | Investig | gational Proc | luct Accountability | 63 |
| | 9.5.1 | Return and | Disposition of Clinical Supplies | 63 |
| 9.6 | Dietary | or Other Pr | otocol Restrictions | 63 |
| 9.7 | Efficacy | y and Safety | Variables | 64 |
| | 9.7.1 | Efficacy ar | nd Safety Measurements Assessed | 64 |
| | 9.7.2 | Efficacy V | ariable | 65 |
| | 9.7.3 | Pharmacok | inetic Variables | 65 |
| | 9.7.4 | Explorator | y Efficacy Variable | 66 |
| | 9.7.5 | Safety Var | iables | 66 |
| | 9.7.6 | Clinical La | boratory Assessments | 67 |
| | 9.7.7 | Explorator | y Sample Analyses | 69 |
| 10 REPC | ORTING | 6 ADVERS | E EVENTS | 70 |
| 10.1 | Adverse | e Events | | 70 |
| 10.2 | Serious | Adverse Ev | vents | 73 |
| 10.3 | Adverse | e Events Oc | curring Secondary to Other Events | 74 |
| 10.4 | Persiste | nt or Recuri | rent Adverse Events | 74 |
| 10.5 | Abnorn | nal Laborato | ry Values | 74 |

| <b>B</b> OMARIN | PAL-003 A8 | Page 19 |
|--------------------------|--------------------------------------|-----------|
| 10.6 Pre-existing Condi | tions | 75 |
| _ | Examination Findings | |
| | rolonged Hospitalization, or Surgery | |
| | ects after Adverse Events | |
| | se Events | |
| | asures | |
| | covigilance Contact Information | |
| | OF MEASUREMENTS | |
| 11.1 Safety and Pharma | cokinetics | 79 |
| | S | |
| 12.1 Prestudy | | 80 |
| 12.2 Screening Visit | | 80 |
| 12.3 Treatment Period | | 80 |
| 12.3.1 Day 1 (W | eek 1) | 81 |
| 12.3.2 Weekly T | elephone Visit | 81 |
| 12.3.3 Substudy | Visits | 82 |
| 12.3.4 Every 8 W | /eeks | 82 |
| 12.3.5 Unschedu | led Hypersensitivity Reaction Visit | 83 |
| 12.4 Study Completion | Early Termination Visit | 83 |
| 13 DATA QUALITY ASS | URANCE | 85 |
| 14 STATISTICAL METHO | ODS AND DETERMINATION OF SAME | LE SIZE86 |
| 14.1 Statistical and Ana | llytical Plans | 86 |
| 14.2 Safety Analysis | | 86 |
| 14.3 Pharmacokinetic A | Analysis | 86 |
| 14.3.1 Pharmaco | kinetic Substudy Analysis | 87 |
| 14.4 Efficacy Analysis | | 87 |
| 14.5 Determination of S | Sample Size | 87 |

| E | BOMARIN | PAL-003 A8 | Page 20 |
|---|---|---|---|
| | 14.6 Handling of Missing | Data | 87 |
| | • | luct of the Study or Planned Analyses | |
| 15 | | OMMITTEE (DMC) | |
| | | JRANCE, AND INDEMNITY | |
| | | AND SOURCE DOCUMENTS | |
| 18 | STUDY MONITORING | AND AUDITING | 92 |
| 19 | RETENTION OF RECOR | RDS | 93 |
| | | I AND PUBLICATION | |
| 21 | REFERENCES | | 95 |
| 22 | INVESTIGATOR RESPO | ONSIBILITIES | 97 |
| | 22.1 Conduct of Study an | d Protection of Human Subjects | 97 |
| 23 | | | |
| 24 | PROTOCOL AMENDME | ENT TEXT REVISIONS | 99 |
| LI | ST OF TABLES | | |
| Tal | ble 9.1.1: Schedule of Ever | nts | 43 |
| Ta | ble 9.1.2: PK Substudy Do | sing Regimens | 46 |
| | | actions in Response to Hypersensitivity A | |
| Tal | ble 9.1.2.1: Brown's Sever | rity Criteria | 50 |
| Ta | ble 9.4.2.1.1: Prefilled Syri | inge Volume, Concentration, and Dose | 57 |
| Tal | ble 9.4.2.1.2: Conversion f | From Vial and Syringe Dose to Prefilled S | yringe Dose58 |
| Ta | ble 9.4.4.1: Fixed Doses fo | or Subjects on Weight-Based Dose Regim | en60 |
| Ta | ble 9.7.1.1: Summary of La | aboratory Assessments | 64 |
| Ta | ble 9.7.6.1: Clinical Labora | atory Tests | 68 |




### 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# Abbreviations

ADR adverse drug reaction

AE adverse event

ALT alanine aminotransferase AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

AUC<sub>0-7 days</sub> area under the plasma concentration-time curve from time zero on Day 1 to Day

8

BUN blood urea nitrogen

°C degree Celsius

C<sub>3</sub> complement 3

C<sub>4</sub> complement 4

CBC complete blood count

CD Compact disk

CFR Code of Federal Regulations
CH50 total hemolytic complement
C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CO<sub>2</sub> carbon dioxide

CRA Clinical Research Associate

CRF case report form
CRP C-reactive protein

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular

DBP diastolic blood pressure
DMC Data Monitoring Committee

ECG electrocardiogram

ETV Early Termination Visit

FDA Food and Drug Administration

F/U follow-up g gram

GCP Good Clinical Practice
GGT gamma-glutamyltransferase

GI gastrointestinal



IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

ID identification

IgEimmunoglobulin EIgGimmunoglobulin GIgMimmunoglobulin MIPinvestigational productIRBInstitutional Review Board

IV intravenous kg kilogram

MedDRA Medical Dictionary for Regulatory Activities

mg milligram mL milliliter

mm Hg millimeter of mercury

NAb neutralizing antibodies

NCI National Cancer Institute

NIAID/FAAN National Institute of Allergy and Infectious Disease/Food Allergy and

Anaphylaxis Network

NOAEL no observable adverse effect level

NSAID non-steroidal anti-inflammatory medication

OTC over the counter

PAH phenylalanine hydroxylase PAL phenylalanine ammonia lyase

PEG polyethylene glycol Phe phenylalanine

PI Principal Investigator
PK pharmacokinetics
PKU phenylketonuria

rAvPAL-PEG recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG

RBC red blood cell

SAE serious adverse event
SAP Statistical Analysis Plan
SBP systolic blood pressure

SC subcutaneous



SD standard deviation SDV source data verified

SGOT serum glutamic oxalo-acetic transaminase SGPT serum glutamic pyruvate transaminase

US United States
WBC white blood cell

# **Definition of Terms:**

# Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use." (from E6 ICH)

The terms "IP" and "study drug" may be used interchangeably in the protocol.



### 5 ETHICS

# 5.1 Institutional Review Board or Ethics Committee

Prior to initiating the study, the Investigator will obtain written confirmation that the Institutional Review Board (IRB) is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, and applicable laws and local regulations. A copy of the confirmation from the IRB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Principal Investigator (PI) will provide the IRB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all consent forms translated to a language other than the native language of the clinical site. The study will not be initiated and investigational product (IP) supplies will not be shipped to the site until appropriate documents from the IRB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the PI and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study were made to the IRB and BioMarin by the PI in accordance with applicable governmental regulations.

# 5.2 Ethical Conduct of Study

This study will be conducted in accordance with the following:

- United States (US) Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- E6 ICH Guideline for GCP
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation; the study will be conducted under a protocol reviewed and approved by an IRB; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each subject, or his or her legally authorized representative will



provide written, informed consent before any study-related tests or evaluations are performed.

# 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, E6 ICH (GCP Guideline, Section 4.8) and 21 CFR Part 50 and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB. BioMarin and the IRB must approve the documents before they are implemented. A copy of the approved ICF, and if applicable, a copy of the approved subject information sheet, minor assent form, parental ICF for studies involving minors, and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or its designee prior to the delivery of study drug.

Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the subject's legally authorized representative) and will maintain the original in the subject's record file.



#### 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

Prior to beginning the study, the PI at each site must provide to BioMarin or its designee a fully executed and signed Form FDA (Food and Drug Administration) 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of research subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin's Pharmacovigilance Department (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required. Some study assessments, including administration of study drug, may be performed at the subject's home. All assessments performed for this study will be administered by clinic staff or other qualified and trained study personnel.

Anti-rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase polyethylene glycol) immunoglobulin E (IgE) antibody analysis will be performed by a vendor; other antibody analysis will be performed by BioMarin. Clinical laboratory tests, including serum pregnancy tests (if applicable), will be analyzed and processed by a central laboratory, with the exception of erythrocyte sedimentation rate (ESR), and urine pregnancy tests (if applicable), which will be analyzed by a local laboratory. A central laboratory will also be used to perform analysis of blood phenylalanine (Phe) concentrations and urinalysis. Pharmacokinetic (PK) analysis will be performed by BioMarin.

Prior to database lock in multicenter studies, a Coordinating Investigator will be identified who will read the clinical study report and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe.



#### 7 INTRODUCTION

A comprehensive review of PEGylated recombinant Anabaena variabilis phenylalanine ammonia lyase (rAvPAL-PEG) is contained in the IB supplied by BioMarin; the Investigator should review this document prior to initiating this study.

# 7.1 Nonclinical Studies

The nonclinical program for rAvPAL-PEG has characterized the pharmacology, pharmacokinetics (PK), and toxicology of rAvPAL-PEG using the intended clinical SC route of administration. Pharmacology was assessed in the BTBR  $Pah^{\rm enu2}$  (ENU2) mouse model of PKU. The ENU2 mouse model exhibits characteristics similar to those of PKU patients, including hyperphenylalaninemia (baseline plasma Phe concentrations of 1000 to 2000  $\mu$ M) and hypopigmentation. Following weekly doses of rAvPAL-PEG administered to male ENU2 mice, plasma Phe concentrations decreased from approximately 2000  $\mu$ M to < 200  $\mu$ M after 2 dose administrations. An attenuated reduction of blood Phe was seen between Week 3 and Week 7 of dosing. After 7 weekly administrations of rAvPAL-PEG, pharmacological activity returned as evidenced by stabilized concentrations of plasma Phe < 200  $\mu$ M over the entire week, which continued for a total of 15 weeks.

In pharmacodynamic studies in the BTBR Pahenu2 (ENU2) mouse model administered 80 mg/kg/week rAvPEG-PAL, two dose interruption assessments were performed: a 2-4 week dose interruption and an 11-week dose interruption. Following both dose interruption assessments, the animals re-started rAvPAL-PEG at a dose of 80 mg/kg/week. No attenuated Phe response was observed when rAvPAL-PEG injections were temporarily stopped for 2-4 weeks, and there was an immediate return to stable blood Phe reductions. A similar interim attenuated response was observed with the longer dose interruption of approximately 11 weeks. In both of these assessments, no safety issues were noted upon re-starting dosing with rAvPAL-PEG (Lapis, 2007, ASHG 57th Annual Meeting).

Safety pharmacology studies were conducted in rats and cynomolgus monkeys. No respiratory or central nervous system (CNS) effects were seen with SC administration of rAvPAL-PEG. No changes in cardiovascular (CV) parameters, including electrocardiogram (ECG) waveforms, were observed in telemetry-instrumented monkeys assessed for the CV effects of rAvPAL-PEG administered subcutaneously.

Pharmacokinetic parameters were evaluated in single-dose and repeat-dose studies in rats and cynomolgus monkeys. The elimination half-life ( $t_{1/2}$ ) values of rAvPAL-PEG administered to normal rats at SC doses of 10, 25, and 250 mg/kg were 47, 33, and 44 hours, respectively,




and exhibited modest area under the plasma concentration-time curve (AUC)-dose. In the cynomolgus monkey after SC administration of rAvPAL-PEG, the  $t_{1/2}$  was 65 hours at 4.0 mg/kg, 71 hours at 12 mg/kg, and could not be determined at 60 mg/kg (the highest dose). Qualitatively, the kinetics of rAvPAL-PEG in the rat and monkey appear to have similar characteristics. The following findings were noted: (1) a 1-compartment model with first-order absorption appears to describe the plasma profiles of rAvPAL-PEG after single-dose administration, (2) absorption is slow and there is a long absorption period after SC administration to maximum observed plasma concentration ( $C_{max}$ ), along with a long  $t_{1/2}$ , (3) elimination is slow and monophasic, (4) there does not appear to be a gender difference, and (5) the AUC and the  $C_{max}$  are roughly linearly proportional.

Toxicology of rAvPAL-PEG was assessed in single-dose and repeat-dose studies in normal rats and cynomolgus monkeys. In the single-dose rat study, decreased body weight gain and Kupffer cell vacuolization at the high SC dose of 250 mg/kg was observed; however, the Kupffer cell finding was not seen in the single-dose study in cynomolgus monkeys. In a 26-week repeat-dose toxicity and toxicokinetic (TK) rat study, decreased body weight gain, decreased food consumption, vacuolation/hypertrophy of the renal tubule cells, and vacuolation of the histiocytic cells were observed in rats administered 25 mg/kg/dose, twice weekly. In a 39-week repeat-dose study in monkeys, arterial inflammation, perivascular cellular infiltrates in the SC injection sites, thymic atrophy, and increased lymphoid nodules in bone marrow of the sternum were observed in monkeys given  $\geq 3$  mg/kg/dose, twice weekly. Of these findings, only the arterial inflammation was deemed adverse and this finding was completely reversed after 13-weeks of recovery. The no-observed-adverse-effect-level (NOAEL) of rAvPAL-PEG when administered subcutaneously twice weekly for 26 weeks and 39 weeks in the rat and monkey, respectively, was 1.0 mg/kg. These NOAELs were based on histological findings of vacuolation/hypertrophy of the renal tubule cells in the rat and arterial inflammation findings in the monkey.

#### 7.2 Previous Clinical Studies

The rAvPAL-PEG clinical development program has been designed to demonstrate the safety and efficacy of rAvPAL-PEG in reducing blood Phe concentrations in PKU subjects who do not respond to treatment with Kuvan® or are not compliant with Kuvan® treatment. This study is an extension of the ongoing human clinical studies with rAvPAL-PEG (Study PAL-002, Study PAL-004, and Study 165-205) based on data from the completed clinical study, PAL-001, and clinical experience from this ongoing study and the other ongoing Phase 2 studies, PAL-002 and PAL-004.



# 7.2.1 Phase 1 Study, PAL-001

The first-in-human trial using rAvPAL-PEG, Study PAL-001, was a Phase 1, open-label, dose-escalation study in PKU subjects in the US. The primary objective was to assess the safety and tolerability of single SC injections of rAvPAL-PEG. Secondary objectives were to evaluate the PK of single, SC injections of rAvPAL-PEG administered at escalating doses in subjects with PKU and to evaluate the effect of rAvPAL-PEG on blood Phe concentrations.

The effectiveness of rAvPAL-PEG in decreasing Phe concentrations in nonclinical studies of ENU2 mice was consistent with what was observed in PAL-001. PAL-001 enrolled 25 PKU subjects with a mean (standard deviation; SD) baseline blood Phe concentration of 1310 µmol/L (405). The 25 subjects who enrolled into the study were assigned to receive a single administration of rAvPAL-PEG at 1 of 5 dose levels: 0.001, 0.003, 0.01, 0.03, and 0.1 mg/kg. Five subjects each received 1 of the 5 dose levels of rAvPAL-PEG.

Key safety, efficacy, and PK results of Study PAL-001 are summarized as follows:

- rAvPAL-PEG was well tolerated and had a clinically significant blood-lowering effect on Phe concentration when administered at a dose of 0.1 mg/kg.
- For the 5 subjects who were administered 0.1 mg/kg rAvPAL-PEG, clinically significant reductions in blood Phe level were observed, with the most clinically significant decreases from baseline values to Day 7, ranging from 33.8% to 97.3% (mean of 58.12%). The mean baseline blood Phe level for these 5 subjects was 1113 µmol/L.
- Overall, no clinically significant reductions in blood Phe level were observed in subjects who were administered rAvPAL-PEG at the lower doses of 0.001, 0.003, 0.01, and 0.03 mg/kg.
- For subjects who were administered rAvPAL-PEG at the 3 higher dose levels
   (0.01, 0.03, and 0.1 mg/kg) and who had measurable rAvPAL-PEG concentration
   levels, the calculated PK parameters were a mean T<sub>max</sub> of 89-106 hours, a t<sub>1/2</sub> of
   46-120 hours, and an AUC<sub>0-t</sub>, and C<sub>max</sub> that were proportional with dose.
   Drug exposure was slightly increased with increased dose.

#### 7.2.2 Phase 2 Studies PAL-002, PAL-004, and 165-205

Based on results from the Phase 1, single-dose study, the Phase 2 studies have been designed to evaluate rAvPAL-PEG at various doses and dosing regimens to safely achieve and maintain blood Phe reductions in subjects with PKU. Currently, there are three ongoing Phase 2 studies (PAL-002, PAL-004, 165-205); an overview of each study is presented in Section 7.2.2.1 (PAL-002), Section 7.2.2.2 (PAL-004), and Section 7.2.2.3 (165-205).




# 7.2.2.1 Study PAL-002

Study PAL-002 (A Phase 2, Open-Label, Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria) was initiated in September 2009 and has completed enrollment. As of 10 September 2012, 40 subjects have been enrolled and 37 have completed the study. PAL-002 enrolled 11 previously exposed subjects from the single-dose study, PAL-001, and 29 subjects who were naïve to rAvPAL-PEG. Thirty-three of the 37 subjects who completed PAL-002 enrolled into this open-label extension study (PAL-003). Two subjects discontinued from the study due to lost to follow-up, relocation, or other reasons, and 1 subject discontinued from the study due to an AE (skin reaction).

The primary objective of this study was to evaluate the effect of multiple doses of rAvPAL-PEG (ranging from 0.001 mg/kg/week to 1.0 mg/kg/week) on blood Phe concentrations in subjects with PKU with up to 16 weeks of treatment. The secondary objectives of the study were to evaluate the safety and tolerability of SC injections of multiple doses of rAvPAL-PEG, to evaluate the immune response to rAvPAL-PEG, and to evaluate the PK profile of rAvPAL-PEG in subjects with PKU.

The PAL-002 study design consists of two parts. In Part 1, rAvPAL-PEG was administered as a once weekly fixed, low-dose induction regimen for 8 weeks. In Part 2, the rAvPAL-PEG dose was titrated upwards; subjects received adjustable dose increases for up to 8 weeks to achieve a target blood Phe concentration of 600 µmol/L. The doses and dosing schedules were revised with a series of protocol amendments to incorporate the information gained during conduct of this early, open-label, multiple-dose study.

A wide range of doses was planned for the PAL-002 study, beginning with doses as low as 0.001 mg/kg/week. However, no substantial reductions in blood Phe level were observed in the majority of subjects who were administered rAvPAL-PEG in the initial four cohorts at doses of  $0.001,\,0.003,\,0.01,\,$  and  $0.03\,$  mg/kg administered once per week. The absence of appreciable Phe reduction after 16 weeks of treatment in this range of doses led to a decision to amend the study protocol to include a cohort with a higher starting dose of  $0.1\,$  mg/kg/week, which had been previously shown to decrease blood Phe levels to approximately  $600\,$  µmol/L in the single-dose, Phase 1 study (PAL-001). After the first 2 weeks of dosing at  $0.1\,$  mg/kg/week, transient Phe reduction was observed in this subset of subjects. However, this dosing regimen was accompanied by mild to moderate hypersensitivity reactions primarily after the second weekly dose, suggesting that additional exploration of dosing regimens would be required.




In summary, preliminary results from PAL-002 demonstrated that doses below 0.1 g/kg administered once per week were not effective in reducing Phe levels. While transient reduction of Phe was apparent at doses of at least 0.1 mg/kg given once per week, this dose regimen was associated with a high incidence of systemic hypersensitivity reactions, typically following the second weekly dose. Further escalation above this dose of 0.1 mg/kg/week would be required to sustain the effect on Phe levels over time. Increased doses would require spreading dose administration over several days per week, as once-weekly administration of higher doses would not be practical due to the large volume of study drug. Therefore, additional dosing regimens would need to be explored in a subsequent study (PAL-004).

Once subjects completed Study PAL-002, they were eligible to enroll into this open-label extension study, PAL-003 to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

# 7.2.2.2 Study PAL-004

PAL-004 (An Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Dose Levels of rAvPAL-PEG Administered Daily in Subjects With Phenylketonuria) was initiated in April 2011 and has completed enrollment. As of 10 September 2012, 16 subjects have been enrolled, 15 subjects have completed the study, and 15 subjects have enrolled into this study (PAL-003). One subject withdrew consent from continued participation prior to study completion. All subjects enrolled in this study were naïve to rAvPAL-PEG exposure.

The objective of this study was to determine if daily administration (defined as 5days/week) of rAvPAL-PEG at dose levels of 0.06, 0.1, 0.2, 0.4, 0.6, and 0.8 mg/kg/day was safe and effective in reducing and maintaining blood Phe concentrations to 600 µmol/L in subjects with PKU. The starting dose was 0.4 mg/kg, administered 5 days/week. A total of 12 subjects were added in sequence and were started on doses of 0.4, 0.2, 0.1, 0.06 mg, or 0.001/kg/day based on incoming safety data. Overall, subjects in PAL-004 who initiated treatment at higher daily doses of 0.1 to 0.4 mg/kg/day achieved immediate and substantial reduction of blood Phe levels, but dosing had to be temporarily reduced or interrupted due to the onset of systemic hypersensitivity reactions at approximately Day 10 of dosing. Phe reductions did not persist in the setting of temporary dose reduction or interruption, but Phe levels generally improved if higher dose levels were reinstated.

To prevent the onset of hypersensitivity reactions that were temporally associated with the onset of anti-drug IgM responses, an additional dosing strategy was assessed in PAL-004;


4 subjects initiated dosing at a low dose of 0.001mg/kg/day or 0.06mg/kg/day for 5 consecutive days and then dosing was suspended for 2 weeks. Dosing was restarted on Day 21 at the initial dose followed by dose titration to target Phe levels. Subjects administered this dosing regimen had similar efficacy, but the incidence of hypersensitivity reactions appeared to be similar to that of subjects who did not have the planned dose interruption, suggesting little advantage with this alternate induction regimen.

Experience from PAL-004 indicated that initiating daily rAvPAL-PEG dosing with relatively high daily doses was not sustainable due to the onset of hypersensitivity reactions that occurred approximately 9 to 12 days after the start of administration, nor was the alternate dosing regimen (2 week drug holiday) well tolerated or effective in Phe reduction. In addition, the daily treatment regimen did not reduce the time to achieve target blood Phe levels seen in previous studies. This study indicated that to improve tolerability, rAvPAL-PEG should be initiated with an induction period at doses substantially lower than 0.4mg/kg, followed by upward dose titration toward target Phe levels.

Once subjects completed Study PAL-004, they were eligible to enroll into this open-label extension study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week.

# 7.2.2.3 Study 165-205

Study 165-205 (A Phase 2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate Safety, Efficacy, and Tolerability of Subcutaneously Administered rAvPAL-PEG in Subjects With PKU for 24 Weeks) was initiated in May 2012. Data from ongoing Studies PAL-002, PAL-004, and PAL-003 suggested that a 4-week treatment course with weekly dosing at a fixed low dose (induction), followed by a weekly 2-fold, upward titration of rAvPAL-PEG to approximately 10-fold higher than the initiation dose (maximum of 375 mg/week) is effective and well tolerated. The objective of this study was to further assess this dosing regimen. Two rAvPAL-PEG dosing regimens were to be explored in this study: weekly low-dose induction (2.5 mg/week for 4 to 8 weeks), followed by a period of upward dose titration towards a target Phe level (600 µmol/L) followed by maintenance dosing at that level through the 24 week study duration (Group 1). The other dosing regimen planned for this study (Group 2) involved administration of a single bolus dose of 8 mg, followed by a treatment holiday of at least 3 weeks duration followed by resumption and escalation of study drug administration following a pattern similar to that employed in Group 1. A total of 24 subjects were enrolled into 165-205. In addition to confirming an effective, well-tolerated dose regimen, this study incorporated non-weight-based dosing, starting with dose



administration once per week at a low dose (2.5mg) with gradual escalation and conversion of dose administration to 5x/week dosing for chronic maintenance therapy.

Once subjects have completed Study 165-205, they are eligible to enroll into this study to continue to receive rAvPAL-PEG up to a maximum dose of 5.0 mg/kg/week or 375 mg/week, or into the Phase 3 study, 165-302.

#### 7.3 Study Rationale

PKU is an autosomal, recessive, inherited disease characterized by deficiency in the enzyme PAH. Approximately 1 in every 10,000 infants in North America is born with PKU (Scriver, 2001, McGraw-Hill). Left untreated, PAH deficiency is associated with an abnormally elevated concentration of Phe, which is toxic to the brain (Kaufman, 1989, J Pediatr.) and can result in a variety of neuropathologic conditions, including mental retardation, microcephaly, delayed speech, seizures, and behavioral abnormalities (Scriver, 2001, McGraw-Hill). The brains of untreated patients with PKU show evidence of hypomyelination and gliosis, arrest in cerebral development, and, in some cases, white matter degeneration (Huttenlocher, 2000, Eur.J Pediatr.). Elevated Phe during fetal development leads to severe mental retardation and can cause microcephaly, growth retardation, and congenital heart disease (Guttler, 2003, Pediatrics), (Koch, 2003, Pediatrics), (Lee, 2003, Pediatrics), (Levy, 2003, Pediatrics), (Matalon, 2003, Pediatrics), (Rouse, 2004, J.Pediatr.).

For a subset of patients with residual enzyme activity, treatment with Kuvan<sup>®</sup> is an option. For all other patients, current management of PKU involves adherence to low-Phe medicinal diet formulas and dietary restriction of Phe-containing foods. Implementation of a Phe-restricted diet in infancy significantly reduces blood Phe concentrations and prevents many of the neuropathologic manifestations of PKU, including severe mental retardation. However, compliance with this restrictive diet can be difficult for older children, adolescents, and adults, and adherence may result in nutritional deficiencies due to the limitations of natural protein sources (Fisch, 2000, Eur.J.Pediatr.), (Walter, 2002, Lancet).

The need exists for a treatment that will help individuals with PKU safely achieve lifelong, reliable control of blood phenylalanine (Phe) concentrations and improve functional outcomes. rAvPAL-PEG is a potential substitute for the phenylalanine hydroxylase (PAH) enzyme, which is defective in individuals with PKU. rAvPAL-PEG may control blood Phe concentrations, which may have additional clinical benefits.

Blood Phe levels depend not only on the functional presence of the endogenous enzyme PAH but also on the dietary intake of Phe. It is important to understand the role of diet on blood Phe levels concurrent with the administration of rAvPAL-PEG treatment. Therefore, an




exploratory objective has been added to this study to assess the relationship of diet, rAvPAL-PEG administration, and blood Phe level. Changes to subject diet are not allowed in this study unless per the Investigator. Diet will be monitored using a diet diary.

A pharmacokinetic (PK) substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Single-dose PK data has been collected in the Phase 1 study, PAL-001. However, there is little multiple-dose PK data or data for when subjects have reached and maintained a stable dosing regimen. With the PK substudy, multiple-dose PK data will be collected for subjects who have already achieved Phe reduction to within the protocol-defined target range.

This study is an extension of previous rAvPAL-PEG Phase 2 studies. Administration of rAvPAL-PEG will be continued to assess the long-term safety and efficacy of rAvPAL-PEG in PKU subjects.

#### 7.4 Summary of Overall Risks and Benefits

It is not expected that data from previous rAvPAL-PEG studies will change the assumption that rAvPAL-PEG has a toxicity profile similar to other recombinant PEGylated non-human enzymes currently in use. The toxicities of these drugs usually fall into 2 main categories: toxicity due to exposure to PEG, and toxicity due to immunologic sensitization. In addition, exaggerated pharmacological effects resulting in very low Phe concentrations could be observed. Other adverse events (AEs) that could occur with rAvPAL-PEG include injection-site reactions and other general symptoms.

#### 7.4.1 Toxicity Due to Exposure to Polyethylene Glycol (PEG)

Acute exposure to high doses of PEG can result in renal toxicity. There have been a few reports of PEG-related AEs in humans; cumulative intravenous (IV) PEG doses of 121 to 240 g caused acute renal tubular necrosis, oliguria, and azotemia. The anticipated PEG exposure associated with the expected rAvPAL-PEG dose range (6 g per week) is at least 80-fold lower than the reported toxic doses and comparable to exposures to PEG in widely used medicines and other compounds that are administered by the IV, oral, rectal, and topical routes (Webster, 2007, Drug Metab Dispos.). No indication of PEG-related toxicity at the ultrastructural level was observed in monkeys given a single dose of up to 60 mg/kg rAvPAL-PEG SC. In rats, both renal tubule vacuolation and histiocytic cell vacuoles have been assocated with PEG-related catabolism and administration of other PEGylated proteins (refer to Section 7.1).




Based on phase 3 data, as of 4MAR2016, there have been no reported events of glomerulonephritis or renal failure reported with pegvaliase administration. Of the 10 subjects identified with UAC ratios  $\geq 3$  mg/mmol on 3 or more consecutive measurements, values were generally in the microalbuminuria range and none had concurrent sustained hematuria. Seven of these 10 subjects had microalbuminuria at baseline prior to pegvaliase exposure, of which 2 events resolved while on pegvaliase treatment and 4 events did not progress while subjects remained on pegvaliase. One of these 7 subjects with baseline microalbuminuria (3.62 mg/mmol at baseline) had an increase in their UAC ratio during the study, which was more apparent after dose titration to 60 mg of pegvaliase (remaining in microalbuminuria range, with a most recent value of 20.36 mg/mmol), however evaluating relationship to pegvaliase treatment is confounded by a medical history of obesity, hypertension, and new onset pre-diabetes during the Phase 3 study that are conditions also associated with development of microalbuminuria. The subject continues on pegvaliase treatment with continued safety monitoring.

Three of the 10 subjects developed new onset microalbuminuria for at least 3 consecutive measurements during the Phase 3 study, one of which resolved while continuing on pegvaliase treatment and 1 subject continues to have fluctuating low level microalbuminuria with intermittent values in the normal range. One subject discontinued from the Phase 3 study after a few intermittent elevations into the microalbuminuria range. The subject had a maximum UAC ratio of 175 mg/g on Day 8 on the study; at the time of study and study drug discontinuation (Day 36), UAC ratio was within the normal range at 19 mg/g. The final study visit recorded for this subject (Day 67) had a UAC ratio of 17 mg/g. This subject reported a single concurrent grade 1 event of urticaria, which resolved in 2 days, and no other reported events suggestive of immune complex disease. None of the subjects described above have developed sustained elevations in serum creatinine or concurrent sustained hematuria.

To monitor for renal toxicity, subjects participating in this study will undergo urinalysis, will be assessed for urine albumin/creatinine ratio, and will undergo blood chemistry tests to assess renal function.

# 7.4.2 Immunologic Response

The active drug substance in rAvPAL-PEG is a bacterial protein and elicits immune recognition and subsequent antibody responses. Antibody epitopes on the protein are expected to be rendered at least partially inaccessible by the extensive PEGylation on the drug (Gamez, 2007, Mol.Genet.Metab). In vivo and in vitro experiments have shown that PEGylation of proteins and cells can attenuate the immunological response (Scott, 1997, Proc.Natl.Acad.Sci.U.S.A), (Chen, 2001, BioDrugs.). PEGylation has been effective in




reducing anti-rAvPAL antibody titers in the mouse model but does not eliminate antibody formation. Although PEGylation of rAvPAL likely reduces the antigenicity of the molecule, 100% of individuals exposed to rAvPAL-PEG develop antibodies against rAvPAL.

Drug-specific immune responses can range from clinical irrelevance to causing serious hypersensitivity AEs (such as anaphylaxis) and may reduce efficacy due to antibody-mediated drug clearance or antibody neutralization of enzymatic activity. Historically, PEG was thought to be nonimmunogenic (Davis, 1981, Clin.Exp.Immunol.), (Harris, 2003, Nat.Rev.Drug Discov.); however, repeated studies have found that subcutaneous (SC) and intravenous exposure to PEG can induce anti-PEG antibodies (Harris, 2003, Nat.Rev.Drug Discov.), (Richter, 1983, Int.Arch.Allergy Appl.Immunol.). In some instances, development of such antibodies did not result in significant clinical effects in humans (Richter, 1984, Int.Arch.Allergy Appl.Immunol.). However, PEG antibody responses were associated with hypersensitivity reactions to PEGylated liposomes (Judge, 2006, Mol.Ther.). Anti-PEG antibodies have also been associated with nonresponsiveness against therapy (Armstrong, 2007, Cancer), (Ganson, 2006, Arthritis Res.Ther.).

Subjects participating in the Phase 2 clinical studies have been monitored closely for anti-drug immunogenicity (anti-rAvPAL immunoglobulin G [IgG], anti-rAvPAL IgM, anti-PEG IgM, anti-PEG IgG, neutralizing antibodies that inhibit PAL enzymatic activity, anti-rAvPAL IgE, and anti-rAvPAL-PEG IgE), complements, C-reactive protein (CRP), ESR, and complete chemistry. All subjects treated with rAvPAL-PEG in the Phase 2 clinical trials developed antibodies against the PAL protein. Anti-rAvPAL IgM antibodies were first detected within 2-3 weeks of treatment initiation and anti-rAvPAL IgG antibodies were detected within 2-3 months. The anti-rAvPAL IgG response generally peaked by 3-5 months and was sustained in all subjects. Neutralizing antibodies (NAb) capable of inhibiting enzymatic activity were detected in a minority of subjects 2-3 months after treatment initiation. The timing of the NAb response suggests these antibodies may be a component of the anti-rAvPAL IgG response. It is expected that the centralized location of the PAL active site, within the tetrameric structure, makes it difficult for antibodies to bind and inhibit enzymatic activity. In addition, anti-PAL antibody binding is likely sterically hindered by the extensive PEGylation. The majority of treated subjects also developed a transient anti-PEG antibody response. The anti-PEG response was comprised of IgM and IgG isotypes. In general, anti-PEG antibodies were no longer detected after 5-6 months of treatment. This type of transient antibody response is typical of T cell-independent type 2 (TI-2) responses.

The majority of immune-mediated AEs experienced in subjects treated with rAvPAL-PEG in the Phase 2 studies are believed to be the result of antibody-mediated hypersensitivity. The




primary immune mediator is thought to be IgM immune complexes, as evidenced by the timing of onset prior to IgG development and the reduced occurrence over time. IgE positive test results have not been associated with hypersensitivity in any of the subjects thus far, and the majority of subjects have been safely rechallenged with rAvPAL-PEG following reactions. IgM immune complexes are known to be efficient activators of the classical complement pathway and can lead to the accumulation of complement component anaphylatoxins (C3a, C4a, C5a) that can induce hypersensitivity symptoms. Although IgG immune complexes can also activate the classical complement pathway, they do so with less efficiency than IgM. This is due, in part, to the requirement for multiple Fc regions in close proximity to activate the complement cascade, meaning that multiple monomeric IgG Abs are required to bind, whereas only one pentameric IgM Ab is needed to bind to activate complement. Also, in the case of rAvPAL-PEG, binding of anti-PAL IgG antibodies is likely compromised due to epitope masking by the PEGylation, which may reduce IgG-mediated complement activation in vivo. This complex dynamic between combined isotype-specific Ab responses and epitope accessibility is thought to be a major factor dictating the need for an induction and titration dose regimen in the treatment of rAvPAL-PEG to be implemented in this study.

## 7.4.3 Management of Hypersensitivity Reactions

Hypersensitivity reactions to the SC injection of rAvPAL-PEG may be mild, moderate, or severe in intensity. Reactions may include pruritus, rash, shortness of breath, hypotension, or anaphylaxis. Clinical assessments should be conducted for a minimum of 30 minutes post-injection. Longer observations may be required at the discretion of the PI. The responsible physician should use all appropriate measures for the treatment of hypersensitivity reactions. Because of the potential for anaphylaxis, equipment for emergency resuscitation (including epinephrine) should be within easy access during and after the rAvPAL-PEG injection. Subject should be pre-medicated with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. If non-steroidal anti-inflammatory medication (NSAIDs) is administered as a premedication, it should be given with food. Subjects who qualify for self-administration of study drug are trained to recognize a serious hypersensitivity AEs and how to respond. Additionally, subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (Section 9.4). Refer to Section 9.1.1.3 for instructions regarding resumption of study drug following resolution of symptoms consistent with a clinical diagnosis of anaphylaxis per National Institute of Allergy and Infectious



Disease/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria (Sampson, 2006, J.Allergy Clin.Immunol.).

In the event of a hypersensitivity reaction, subjects may be asked to see an allergist/immunologist and/or provide up to 3 additional blood samples for immunology studies and complement testing. This additional testing may occur up to 6 months following the final study visit.

The following measures are recommended for the treatment of hypersensitivity reaction symptoms:

- Maintain the airway.
- Vital sign check.
- Administration of oral or IV diphenhydramine.
- Administration of epinephrine if appropriate.
- Administration of oral or IV glucocorticoids.
- Administration of oxygen and IV fluids.
- Administration of additional symptomatic treatment.
- Transfer to an acute care facility of the study center.

In addition, clinical judgment must be used in determining the appropriateness of corticosteroid administration. An allergy and/or immunology consultation should be sought if necessary. Detailed instructions for the management of hypersensitivity reactions are provided in the Study Reference Manual.



#### 8 STUDY OBJECTIVES

The primary objective of the study is:

• To evaluate the effect of long-term administration of multiple doses of SC injections of rAvPAL-PEG on blood Phe concentrations in subjects with PKU.

The secondary objectives of the study are:

- To evaluate the safety and tolerability of long-term administration of subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU.
- To evaluate the immune response to long-term administration of SC injections of rAvPAL-PEG in subjects with PKU.

The exploratory objective of the study is as follows:

• To evaluate the long-term relationship of diet and change in blood Phe concentration following administration with rAvPAL-PEG in subjects with PKU.

The Substudy objective is as follows:

• To evaluate steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe concentration and for whom no further dose modifications are planned.



#### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a long-term extension of rAvPAL-PEG Phase 2 studies in up to 100 subjects with PKU. The doses are planned to be in the same range as those previously tested in the Phase 2 studies (starting at 0.001 through 5.0 mg/kg/week or 2.5 mg through 375 mg/week), provided no dose-limiting toxicity was observed in a previous rAvPAL-PEG studies. Subjects' doses will not exceed 375 mg/week.

Only subjects who completed a previous rAvPAL-PEG study will be enrolled into this study. Subjects enrolling into PAL-003 with no interruption in dosing from a previous rAvPAL-PEG study may either continue their previous dosing regimen or begin this study at a higher dose level. Subjects who have had dosing interruptions between the previous rAvPAL-PEG study and PAL-003 must have their starting dose determined per the sponsor's medical monitor. The first week of dosing will be administered in the clinic, and the subject must be observed for 30 minutes following administration. Subjects are given two epinephrine injectors and are instructed to carry one epinephrine injector with them at all times (refer to Section 9.4). A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing.

Diet should not be altered during the course of this study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. To monitor for changes in subject diet, a diet diary will be issued to subjects for completion and will be brought to clinic monthly for review with the clinical study staff.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects must meet a set of criteria to be considered appropriate for self-administration. Refer to Section 9.4 for the criteria for which subjects may qualify for self-administration. Additional information is provided in the Subject Self-Administration Training Materials. Additional training will be provided and demonstration of competency required when prefilled syringe drug product is introduced, every 24 weeks, and more often as needed.

Subjects will be evaluated for safety throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.



In addition to the Sponsor, a Data Monitoring Committee (DMC) will monitor the safety of subjects in the study. The DMC is an independent committee that will act in an advisory capacity to the Sponsor.

PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects' previous rAvPAL-PEG dosing will generally continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attempt to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose. Doses will be evaluated on an individual basis.

Evaluations, observations, and procedures will be conducted at selected time points as shown in Table 9.1.1 and Table 9.1.2. After the subject's blood Phe concentration has been controlled to within a target range (60-600  $\mu$ mol/L), the subject may be asked to have additional blood draws for PK and blood Phe concentration analyses as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

A subject will continue in PAL-003 until one of the following occurs:

- The subject withdraws consent and discontinues from the study.
- The subject is discontinued from the study at the discretion of the Investigator or Sponsor.
- The subject has completed the study through the Week 476 visit.
- The study is terminated.
- The study drug receives marketing authorization.

Because the risks of taking BMN 165 during pregnancy and breastfeeding are unknown, subjects cannot take BMN 165 if they are trying to conceive, are pregnant, or are breastfeeding (refer to Section 9.3.2 for Exclusion Criteria). Male subjects who are planning to impregnate a female partner and female subjects who are trying to become pregnant during the study must be temporarily discontinued from study drug for 4 weeks prior to trying to conceive. During that time, subjects must use two acceptable methods of contraception. Subjects who are planning to become pregnant (or impregnate a female partner) may modify their diet in consultation with the investigator and/or study dietician. Subjects who are confirmed to be pregnant per a serum pregnancy test and are temporarily off study drug are not required to perform the scheduled urine pregnancy tests. Subjects who are pregnant or are trying to conceive and have temporarily discontinued study drug should not perform the scheduled PK assessments. Male subjects who have impregnated a female partner may




re-start study drug after conception following the investigator's consultation with and approval by the medical monitor. Male subjects must return to the study-required contraception use (refer to Section 9.3.1 for Inclusion Criteria), which must include one barrier method, prior to restarting study drug. Female subjects who remain in the study after temporary discontinuation of study drug due to pregnancy may restart BMN 165 dosing after a confirmed negative urine pregnancy test result, the birth has been reported (or termination of the pregnancy), and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to conceive. Re-starting BMN 165 dosing requires the investigator's prior consultation with and approval by the medical monitor. Female subjects must return to the study-required contraception use (refer to Section 9.3.1), which must include one barrier method, immediately after the birth (or termination of the pregnancy).

Subjects may withdraw from treatment with study drug at any time; however, subjects will be asked to continue to perform the study assessments until study completion. Subjects may also withdraw from study participation at any time. Because the completeness of the data affects the integrity, accuracy, and interpretation of study results, every effort should be made to retain subjects in the study and to have them complete the study assessments as scheduled as long as continued participation does not compromise subject safety.

A PK substudy has been added to evaluate the steady-state PK of rAvPAL-PEG in up to 6 subjects who have achieved and maintained target blood Phe for at least 2 consecutive measurements and for whom no further dose modifications are planned. Subjects enrolled into the substudy will have additional pre-dose PK sampling performed (refer to Table 9.1.2).

The Schedule of Events and PK substudy collection schedules are presented below in Table 9.1.1 and Table 9.1.2.

| B <b>!</b> OMARIN | PAL-003 A8 | Page 43 |
|-------------------|------------|---------|
|-------------------|------------|---------|

**Table 9.1.1: Schedule of Events** 

| | | Treatment Po | | d <sup>b,c</sup> | | | |
|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Every 8 Weeks <sup>b</sup> | Self-<br>Administration | Study<br>Completion/Early<br>Term. Visit | Unsched. Hyper.<br>Reaction Visit. <sup>d</sup> |
| Assessments and<br>Events | Screening <sup>a</sup> | D 1 | Starting at Week | | | 4 weeks after final dose | Perform within 24 hours |
| Informed consent | X | <i>D</i> 1 | - | | | uose | 2 i nours |
| Medical history, including | | | | | | | |
| allergy history, and | X | | | | | | |
| demographics | | | | | | | |
| Physical examination <sup>e</sup> | X | X | | X | | X | |
| Vital signs <sup>e</sup> | X | X | | X | | X | X |
| Weight | X | | | X | | | |
| 12-lead ECG | X | | | | | X | |
| Clinical laboratory tests <sup>f</sup> | X | | | X | | X | $X^g$ |
| Complements C <sub>3</sub> and C <sub>4</sub> <sup>h</sup> | X | | | X | | | $X^g$ |
| Sedimentation rate | | X | | X | | X | |
| Chest x-ray | X | | | X<br>(Week 48 visit<br>only) | | X | |
| Urine pregnancy test <sup>i</sup> | X | X | | X | | X | |
| Adverse events <sup>j,k</sup> | X | X | X | X | X | X | X |
| Weekly phone call to self admin<br>participants only (to assess AEs,<br>Inj site reactions, concomitant<br>medications) | | | X | | X | | |
| Concomitant medications | X | X | X | X | X | X | X |
| Diet query | X | X | | X | | X | |
| 3-Day diet diary <sup>l</sup> | | | | X | | X | |
| Serum antibodies <sup>m</sup> | | X | | X | | X | X |
| Plasma Phe and plasma<br>tyrosine <sup>n</sup> | X | X | | X <sup>m</sup> | | X | |

|----------|------------|---------|
|----------|------------|---------|

| | | | Treatment Period <sup>b</sup> | o,c | | | |
|---|---|---|---|---|---|---|---|
| | | Week 1 | Weekly<br>Telephone<br>Contacts | Every 8 Weeks <sup>b</sup> | Self-<br>Administration | Study<br>Completion/Early<br>Term. Visit | Unsched. Hyper.<br>Reaction Visit. <sup>d</sup> |
| Assessments and | | | Starting at Week | | | 4 weeks after final | Perform within |
| Events | Screeninga | D 1 | 2 | | | dose | 24 hours |
| Urine albumin/creatinine ratio ° | | | | | | | X |
| Urine N-methyl histamine | | | | | | | X |
| Plasma PK sample <sup>p</sup> | | X | | X | | X | |
| Administer study drug <sup>q</sup> | | X | | X | X | | |
| Training (prefilled syringe) <sup>r</sup> | | | | X<br>Every 24 weeks<br>only | | | |
| Skin biopsy (optional; affected and not affected area) | | | | | | | X |
| Serum tryptase level <sup>s</sup> | | | | | | | X |

AE, adverse event; C<sub>3</sub>, complement 3; C<sub>4</sub>, complement 4; CH50, total hemolytic complement; CRP, C-reactive protein; D, day; ECG, electrocardiogram; eCRF, electronic Case Report Form; ETV, Early Termination Visit; F/U, Follow-up; Hyper, hypersensitivity; IgE, immunoglobulin E; IgG, immunoglobulin G; IgM, immunoglobulin M; IP, investigational product; PK, pharmacokinetics; Phe, phenylalanine; SAE, serious adverse event; Wk, week.

<sup>&</sup>lt;sup>a</sup> A separate Screening visit for this study is required only if the time between completion of the previous rAvPAL-PEG study and enrollment into PAL-003 is greater than 28 days.

<sup>&</sup>lt;sup>b</sup> Visits must be performed in the clinic.

<sup>&</sup>lt;sup>c</sup> On days that a dose is given, all procedures should be performed predose, except where noted.

<sup>&</sup>lt;sup>d</sup> Refer to Section 9.1.1 and Section 12.3.6.

<sup>&</sup>lt;sup>e</sup> Complete physical examinations to include the evaluation of all major body systems. Height will be measured at Screening only.

<sup>&</sup>lt;sup>f</sup> Clinical laboratory tests to include spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis. Urine microscopy will be performed if any urinalysis results are positive for hematuria. It is recommended that urine samples are obtained as a first or second morning void. In the event of elevated urinary protein on a test result, a repeat urinalysis should be performed. This repeat urine sample must be performed in the morning at the first or second morning void to allow for accurate test results and may be performed by a home healthcare nurse. Refer to Table 9.7.6.1.

g Subjects who have a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade ≥ 3 hypersensitivity AE should be assessed for CRP, CH50, C1, C3, and C4 within 24 hours of the reaction.

|----------|------------|---------|
|----------|------------|---------|

- <sup>h</sup> Complement C3 and C4 will be collected at the Screening Visit and every 8 weeks. Additional complement testing may be performed as needed to resolve previous abnormal test results.
- <sup>1</sup> If positive or equivocal, perform serum pregnancy test. Subjects who are confirmed to be pregnant per a serum pregnancy test and are temporarily off study drug are not required to perform the scheduled urine pregnancy tests. Subjects who are planning to become pregnant (or impregnate a female partner) may modify their diet in consultation with the investigator and/or study dietician. Also refer to Section 9.1.
- <sup>j</sup> If any injection site reaction is observed, the corresponding adverse event data must specify injection location (identify current vs. previous visit's injection, eg, right arm vs. left arm). If there is a skin reaction that lasts ≥ 14 days, the Skin Reaction eCRF should be completed. Subjects who experience an injection-site skin reaction that lasts ≥ 14 days should be referred to a dermatologist for consultation and a skin biopsy. It is recommended that a photograph of the skin reaction be taken by the subject or the site to help assess the event; photographs may be collected by the sponsor.
- <sup>k</sup> The reporting period for SAEs begins when informed consent is obtained and continues through 4 weeks after last dose or completion of study participation, whichever occurs last. The reporting period for nonserious AEs is from the first administration of study drug through 4 weeks after last dose or the Study Completion Visit/Early Termination Visit, whichever occurs last. The reporting period for device-related events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe.
- <sup>1</sup> It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.
- <sup>m</sup> For unscheduled hypersensitivity reaction visit, draw serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only; sampling must be performed > 8 hours after event onset and before the next dose of study drug.
- <sup>n</sup> Samples should be drawn at least 2.5 hours after a meal. At the Investigator's discretion, blood Phe may be collected more often should more frequent monitoring of blood Phe levels be clinically warranted.
- $^{\circ}$  It is recommended that urine samples are obtained as a first or second morning void. Subjects with a confirmed urine/albumin creatinine ratio of  $\geq 100$  mg/g should be referred to a nephrologist for consultation if results were within normal range at baseline. Subjects who had elevated results at baseline followed by a confirmed subsequent increase of 100-200 mg/g from baseline should also be referred to a nephrologist for consultation.
- <sup>po</sup> Sampling should be performed predose. Subjects who are pregnant or are trying to conceive and have temporarily discontinued study drug should not perform the scheduled PK assessments.
- <sup>q</sup> Dosing is up to 5.0 mg/kg/week or 375 mg/week, including subjects who receive more than 1 dose/week. Every effort should be made to adhere to the study drug administration regimen. If a subject misses more than 2 scheduled doses of study drug, both dose level and dose frequency may be re-evaluated.
- <sup>r</sup> Initial training on the use of prefilled syringe occurs at the next monthly visit and each subsequent day after transition until (in clinic or by HHRN) it has been determined the subject will switch to prefilled syringe. Once competency is documented, subjects can self-administer study drug using the prefilled syringe. Regular refresher prefilled syringe training occurs in the study clinic every 24 weeks thereafter.
- <sup>s</sup> Mandatory for subjects who have a hypersensitivity AE. Perform within 24 hours of event onset.

| B <b>!</b> OMARIN | PAL-003 A8 | Page 46 |
|-------------------|------------|---------|
|-------------------|------------|---------|

**Table 9.1.2: PK Substudy Dosing Regimens** 

| Treatment Frequency | Plasma PK Sampling | Example |
|---|---|---|
| Subjects who are<br>administered study drug<br>once per week | Pre-dose and every 24 hours<br>thereafter (24, 48, 72, and 96 hours<br>when possible), and pre-dose of the<br>next weekly dose | If dosed on Monday: Obtain PK sample pre-dose when possible – pre-dose Monday, Tuesday, Wednesday, Thursday, Friday, and pre-dose the following Monday. No further PK substudy draws. |
| Subjects who are administered study drug two or three times per week | Pre-dose and every 24 hours during the longest period between doses, when possible, and pre-dose of the next dose. | If dosed on Monday, Thursday, and Friday: Obtain PK sample every 24 hours during the longest period between doses: Pre-dose Monday, Tuesday, Wednesday, and pre-dose Thursday. No further PK substudy draws. |
| Subjects who are administered study drug four to seven times per week. | Pre-dose and every 12 hours during<br>the longest period between doses,<br>when possible, then pre-dose of the<br>next dose. | If dosed Monday through Friday: Obtain PK sample every 12 hours during the longest period between doses (Friday to Monday): pre-dose Friday, 12 hours post-dose Friday, Saturday (24 and 36 hours post dose), Sunday (48 and 60 hours post-dose), and pre-dose the following Monday. No further PK substudy draws. |



#### 9.1.1 Response to Hypersensitivity Adverse Events

Subjects are evaluated for safety throughout the study and are trained to recognize potential hypersensitivity AEs (including anaphylaxis) and how to respond. Subjects are instructed to contact the investigator for any suspected hypersensitivity AE. The investigator may require further evaluation at the clinic. If a hypersensitivity AE (eg, injection-site reaction, rash, joint pain, itching) occurs, the subject may be advised to premedicate with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to subsequent rAvPAL-PEG doses. If NSAIDs are administered as a premedication, they should be given with food. Subjects who experience an injection-site skin reaction that lasts ≥14 days should be referred to a dermatologist for consultation and a skin biopsy.

Hypersensitivity AEs, including anaphylaxis, are expected with rAvPAL-PEG administration. rAvPAL-PEG dosing in response to a suspected hypersensitivity AE may be modified or halted depending on the severity of the event and suspected rAvPAL-PEG causality (Section 9.1.1.3). Severity for hypersensitivity AEs will be per NCI-CTCAE grades.

## 9.1.1.1 Individual Stopping Criteria

Subjects who have an NCI CTCAE grade  $\geq 3$  hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor may be permanently discontinued from study drug.

# 9.1.1.2 Dosing in Response to Hypersensitivity Adverse Events

Dosing in response to a hypersensitivity AE depends on the NCI-CTCAE grade and suspected relationship to rAvPAL-PEG. Dosing instructions are presented in Table 9.1.1.2.1 and are regardless of previous occurrence:

|----------|------------|---------|
|----------|------------|---------|

Table 9.1.1.2.1: Dosing Instructions in Response to Hypersensitivity Adverse Events

| NCI-CTCAE<br>Grade <sup>a</sup> | Related to<br>Study Drug | Actior<br>Maintain <sup>b</sup> | n with Study<br>Reduce <sup>c</sup> | Drug Interrupt <sup>c</sup> | Individual<br>Stopping<br>Criteria <sup>d</sup> | HRV<br>Assessment <sup>e</sup> |
|---|---|---|---|---|---|---|
| 1 | Yes or No | X | (X)<br>Optional | (X)<br>Optional | Cincina | Investigator discretion |
| 2 | Yes or No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 3 | No | X | (X)<br>Optional | (X)<br>Optional | | Investigator discretion |
| 3 | Yes | X | (X)<br>Optional | (X)<br>Optional | | Yes |
| and is suspected to<br>meet Brown's<br>criteria for severe d | Yes | | | | X<br>Consult with<br>sponsor medical<br>monitor | Yes |
| 4 <sup>d</sup> | Yes or No | | | | X<br>Consult with<br>sponsor medical<br>monitor | Yes |

AE, adverse event; CTCAE, Common Terminology Criteria for Adverse Events, version 4.03; HRV, Hypersensitivity Reaction Visit; NCI, National Cancer Institute.

#### 9.1.1.3 Response to Anaphylaxis

If the investigator suspects that the event is anaphylaxis, the subject will be assessed in the clinic. Laboratory assessments for suspected anaphylaxis events should be performed prior to the next administration of study drug (if applicable) and include anti-rAvPAL IgE and

<sup>&</sup>lt;sup>a</sup> NCI-CTCAE grade determination is performed by the investigator and may be done either via telephone or clinic visit.

<sup>&</sup>lt;sup>b</sup> The investigator will instruct the subject to maintain the rAvPAL-PEG dose at the time of AE onset until improvement to grade 1 or resolution (per investigator assessment in the clinic or via telephone).

<sup>&</sup>lt;sup>c</sup>The rAvPAL-PEG dose may be reduced or interrupted if necessary per investigator determination.

<sup>&</sup>lt;sup>d</sup> If a subject has an NCI-CTCAE grade ≥3 hypersensitivity AE that is related to study drug and is suspected to meet Brown's criteria for severe (grade 3) in the judgment of the investigator and the sponsor's medical monitor, the subject may be permanently discontinued from study drug.

<sup>&</sup>lt;sup>e</sup> If the investigator determines that the NCI-CTCAE grade ≥3 hypersensitivity AE is related to administration with rAvPAL-PEG, the subject will be asked to return to the clinic within 24 hours of event onset for evaluation, including laboratory tests (chemistry, hematology, urinalysis, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE [sampling must be performed >8 hours after event onset and before the next dose of study drug], urine albumin/creatinine ratio, urinary N-methyl histamine, CRP, C3, C4, and tryptase).



anti-rAvPAL-PEG IgE (sampling must be performed >8 hours after event onset and before the next dose of study drug) and tryptase (within 24 hours of event onset). The investigator will consult with the sponsor's medical monitor, and a decision will then be made whether to discontinue the subject from study drug, restart dosing at the same dose level, or restart dosing at a lower dose level.

For the first week of dosing after resolution of anaphylaxis, the study drug will be administered in a clinic setting with equipment for emergency resuscitation (including epinephrine) within easy access. The subject must be observed for 30 minutes following administration due to restarting dosing. Additionally, the subject should be premedicated with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to each dose of study drug for one week upon return to dosing regardless of the duration of dose interruption. If NSAIDs are administered as a premedication, they should be given with food.

## 9.1.2 Study Stopping Criteria

If an NCI-CTCAE grade  $\geq$  3 hypersensitivity treatment-related event occurs and meets Brown's criteria for severe (grade 3), an ad hoc independent DMC meeting will convene within 7 days of the event to review and advise the sponsor on potential changes to the study conduct. Clinically severe hypersensitivity is defined as significant hypoxia, hypotension or neurologic compromise that is life-threatening or required treatment to prevent a life-threatening event:

- Cyanosis or  $SpO_2 \le 92\%$
- Hypotension with SBP < 90 mm Hg (adults)
- Neurologic alteration: loss of consciousness, collapse, incontinence

Brown's severity criteria are presented in Table 9.1.2.1.

|----------|------------|---------|
|----------|------------|---------|

Table 9.1.2.1: Brown's Severity Criteria

| Brown's Criteria for<br>Hypersensitivity Reactions | Definition |
|---|---|
| Mild (1) skin and subcutaneous tissue | Generalized erythema, urticaria, periorbital edema, or angioedema |
| Moderate (2) features suggested respiratory, cardiovascular, or gastrointestinal involvement | Dyspnea, stridor, wheeze, nausea, vomiting, dizziness (pre-syncope), diaphoresis, chest or throat tightness, or abdominal pain |
| Severe (3) hypoxia or neurologic compromise | Cyanosis or $SpO_2 \le 92\%$ at any stage, hypotension (SBP < 90 mm Hg in adults), confusion, collapse, loss of consciousness, or incontinence |

#### 9.1.3 Dose Modifications

## 9.1.3.1 Dose Increase Methodology

Each subject's dose may be modified based on the decision of the Investigator. Decisions regarding dose increases will depend on a subject's adverse event profile and blood Phe and drug concentrations.

An individual subject's dose may be adjusted beginning on Day 1 of PAL-003. For the duration of this study, an individual subject's dose may be adjusted if warranted per a subject's adverse event profile and blood Phe concentrations. Dose increases should be performed as follows:

- The dose may be increased by increments of no more than 10-fold higher than the subject's current dose.
- When increasing the dose, a dose may be used that is between the dose levels (0.001, 0.003, 0.01, 0.03, 0.06, 0.1, 0.2, 0.3, 0.4, 0.6, 0.8, 1.0, 2.0, 3.0, 4.0, and 5.0 mg/kg or 2.5, 5, 10, 20, 40, 75, 150, 225, 300, 375 mg/week) or per Investigator determination based on available information regarding a subject's blood Phe (60-600 μmol/L) as well as any adverse events for an individual subject. Dose increases >350 mg/week require consultation with the sponsor's medical monitor.
- The dose may be adjusted by increasing the frequency up to daily-for a total weekly dose not to exceed 5.0 mg/kg or 375 mg/week. Dose increases > 350 mg/week require consultation with the sponsor's medical monitor.
- When a dose is increased, the subject must be observed for 30 minutes following the first modified dose administration. Subjects who increase their dose frequency do not need to be observed following injection of study drug if the increase in frequency does not increase the overall weekly dose amount.
- Only 1 dose adjustment is allowed every 2 weeks.



# 9.1.3.2 Dose Decrease Methodology

Decisions regarding dose decreases will depend on available information regarding a subject's blood Phe (60-600  $\mu$ mol/L), as well as any adverse event (any hypersensitivity reaction as defined in Section 9.1.1). Dose decreases may occur for hypophenylalanemia or any adverse event that may be improved with a lower dose.

A dose should first be reduced by dose level (5.0, 4.0, 3.0, 2.0, 1.0, 0.8, 0.6, 0.4, 0.3, 0.2, 0.1, 0.06, 0.03, 0.01, 0.003, 0.001 mg/kg or 375, 300, 225, 150, 75, 40, 20, 10, 5, and 2.5 mg/week). It is also permitted to decrease dose in between these specified dose levels. If further dosing adjustments are required in response to safety, dosing frequency may also be adjusted.

If the subject develops low blood Phe (as defined by a blood Phe level  $\leq$  30  $\mu$ mol/L ), the subject's rAvPAL-PEG dose should be decreased to the next lower dose. If the condition persists after another 1 month at the lower dose, the dose should be decreased again to the next lower level. If the subject continues to experience low blood Phe after two dose level reductions, the subject may be asked to consult the dietician to eliminate medical foods and/or formulas and to ensure a balanced and nutritious diet (as part of the routine standard of care for PKU disease management, subject diet should be monitored by a dietician).

# 9.2 Discussion of Study Design, Including Choice of Control Group

This open-label, Phase 2 trial was designed to be closely monitored with the goal of obtaining information about the efficacy, safety, tolerability, and PK of long-term administration of rAvPAL-PEG in subjects with PKU. There will be no control group in this study.

#### 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- 1. Must have completed participation in a previous rAvPAL-PEG study.
- 2. Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
- 3. Willing and able to comply with all study procedures.

|----------|------------|---------|
|----------|------------|---------|

- 4. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
- 5. Sexually active subjects must be willing to use two acceptable methods of contraception while participating in the study. Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
- 6. Maintained a stable diet.
- 7. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

#### 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- 1. Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
- 2. Use of any medication other than rAvPAL-PEG that is intended to treat PKU within 14 days prior to the administration of study drug.
- 3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 6 months prior to Screening and during study participation.
- 4. A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product. Subjects with a prior systemic reaction may be eligible for participation per the discretion of the Principal Investigator in consultation with the sponsor's medical monitor. However, subjects who discontinued from study drug early due to a reaction are not eligible to enroll into this study.
- 5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
- 6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).



- 7. Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
- 8. Known hypersensitivity to rAvPAL-PEG necessitating early termination from a previous rAvPAL-PEG study or known hypersensitivity to any of its excipients.
- 9. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
- 10. Creatinine > 1.5 times the upper limit of normal.

# 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representative) may withdraw their consent to participate in the study or to receive study drug at any time without prejudice. The Investigator must withdraw from the study or study drug treatment any subject who requests to be withdrawn. A subject's participation in the study may be discontinued at any time at the discretion of the Investigator and in accordance with his/her clinical judgment. When possible, a subject who is discontinued from study drug should continue to perform the study tests and evaluations until study completion. For subjects who discontinue from the study, the tests and evaluations listed for the Early Termination Visit should be carried out (refer to Section 12.4).

BioMarin must be notified of all subject withdrawals as soon as possible. BioMarin also reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation by an individual Investigator or site for poor enrollment or noncompliance.

Reasons for which the Investigator or BioMarin may withdraw a subject from the study drug include, but are not limited to, the following:

- Subject experiences a serious or intolerable adverse event (AE).
- Subject develops a clinically significant laboratory abnormality.
- Subject requires medication prohibited by the protocol.
- Subject becomes pregnant (refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy and refer to Section 9.1 for details on re-introduction of study drug following pregnancy and breastfeeding).

Reasons for which the Investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject does not adhere to study requirements specified in the protocol.
- Subject was erroneously admitted into the study or does not meet entry criteria.
- Subject is lost to follow-up.



If a subject fails to return for scheduled visits, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone within 7 days, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting contact with the Investigator. This information should be recorded in the study records.

The Investigator or designee must explain to each subject, before enrollment into the study, that for evaluation of study results, the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB. It is the Investigator's (or designee's) responsibility to obtain written permission to use protected health information per country-specific regulations, such as the Health Insurance Portability and Accountability Act (HIPAA) in the United States, from each subject, or if appropriate, the subject's legally authorized representative. If permission to use protected health information is withdrawn, it is the Investigator's responsibility to obtain a written request, to ensure that no further data will be collected from the subject and the subject will be removed from the study.

## 9.3.4 Subject Identification and Replacement of Subjects

Subjects will retain the same subject number assigned in their previous rAvPAL-PEG study. This unique identifier will be on all case report form (CRF) pages. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used.

Subjects who do not complete the study will not be replaced.

#### 9.4 Treatments

Upon enrollment into this study, subjects from previous rAvPAL-PEG studies will be dosed with the same or higher dose that was administered upon completion of that study provided that there was no interruption in dosing. rAvPAL-PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be adjusted per Investigator determination based on available information regarding a subject's blood Phe level (60-600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity reaction) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 weeks will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

Subjects may self-administer study drug at home if approved by the Investigator and the sponsor's medical monitor and if adequate training is demonstrated. Subjects may be eligible to self-administer study drug if he or she meets the following criteria:

|----------|------------|---------|
|----------|------------|---------|

- The subject has no cognitive impairments that may increase the safety risk of self-administration per the assessment of the investigator.
- The subject has been approved for self-administration of study drug by the sponsor's medical monitor.
- The subject has completed the Self-Administration Training conducted by qualified study site personnel and has been observed by the study site personnel to be able to adequately prepare the proper dose and perform the injections safely.
- The subject has been provided with two epinephrine injectors and has been trained on when and how to administer it. The subject will be instructed to carry one epinephrine injector with them at all times.

Qualified study site personnel will train each eligible subject on all procedures for self-administration of study drug (vial and syringe and prefilled syringe drug products) under the supervision of the PI. Qualified study site personnel will also be required to observe the subject prepare and perform at least 1 injection prior to allowing the subject to self-administer a dose at home. The subject will see a study site nurse or home healthcare nurse in person every week or receive a telephone call from site staff to ensure that the subject continues to perform all self-administration procedures correctly, to assess adverse events, and to answer questions throughout the duration of the study. The study site nurse or home healthcare nurse will also perform the regularly scheduled assessments and procedures as outlined in Table 9.1.1 and Section 12; the subject must perform a clinic visit monthly at minimum. Training materials and other information specific to the study site personnel are provided in the Subject Self-Administration Training Materials. Prefilled syringes are dispensed to subjects only after the subject (or caregiver) has completed training and competency is demonstrated in the clinic. Additional regular refresher training occurs in the clinic, every 24 weeks, and more often as needed.

Subjects who are eligible for self-administration will be provided with a Subject Study Manual. Self-administration training materials will be provided in the Subject Study Manual to supplement the in-person training provided by the qualified study site personnel. The Subject Study Manual will include step-by-step instruction on the following:

- How to prepare and perform the injections of study drug safely.
- How to receive, track, store, prepare, and return both used and unused study drug.
- How to safely use and dispose of syringes, including prefilled syringes, used for injections of study drug.
- How to use a new syringe and vial or new prefilled syringe every time drug is administered.

|----------|------------|---------|
|----------|------------|---------|

- How to care for their injection site after an injection of study drug.
- How to identify an adverse reaction and how to report this reaction to the study site.
- How and when to use epinephrine injectors.
- Who to contact at the study site in case of an emergency.

The PI or the sponsor's medical monitor may request that self-administration be halted at any time and that the subject resume injections performed by the study site personnel or home healthcare nurse.

Subjects who are within the target Phe range may also be permitted to convert from weight-based dosing to fixed dosing (refer to Section 9.4.4).

#### 9.4.1 Treatments Administered

BioMarin and/or its designee will provide the study site or subject with a supply of IP sufficient for the completion of the study. BioMarin is responsible for shipping study drug to the clinical sites. The clinical site is responsible for supplying the study drug to subjects who qualify for self-administration. Refer to the PAL-003 Pharmacy Manual for information pertaining to the distribution of study drug from sites.

Information regarding supplying study drug to subjects who qualify for self-administration is provided in the Subject Self-Administration Training Materials.

# 9.4.2 Identity of Investigational Product (IP)

#### 9.4.2.1 Product Characteristics and Labeling

The investigational product is rAvPAL-PEG (recombinant Anabaena variabilis phenylalanine ammonia lyase-PEG). rAvPAL-PEG will be provided in vials or prefilled syringes; subjects will be supplied with vials and syringes or prefilled syringes for administration in the clinic and self-administration:

• rAvPAL-PEG will be provided in 3 mL (milliliter) vials, each containing 1.5±0.2 mL to deliver 15 mg of rAvPAL-PEG per 1.0 mL (15 mg/mL protein concentration). Each vial is filled with 1.5 ± 0.2 mL to allow the withdrawal and delivery of up to 1.0 mL of the drug product.

Or

• rAvPAL-PEG will be provided in 3-mL vials, each containing 1.8±0.3 mL to deliver 20 mg of rAvPAL-PEG per 1.3 mL (15 mg/mL protein concentration). Each vial is filled with 1.8±0.3 mL to allow withdrawal and delivery of up to 1.3 mL.

|----------|------------|---------|
|----------|------------|---------|

Or

• rAvPAL-PEG will be provided in prefilled syringes in three sizes that deliver up to 1 mL. Syringe sizes are 2.5 mg (5 mg/mL protein concentration), 10 mg (20 mg/mL protein concentration), and 20 mg (20 mg/mL protein concentration).

Table 9.4.2.1.1: Prefilled Syringe Volume, Concentration, and Dose

| Prefilled Syringe | Volume | Concentration | Dose |
|-------------------|--------|---------------|--------|
| Sku #1 | 0.5 mL | 5 mg/mL | 2.5 mg |
| Sku #2 | 0.5 mL | 20 mg/mL | 10 mg |
| Sku #3 | 1.0 mL | 20 mg/mL | 20 mg |

Subjects who have undergone training and who have demonstrated competency on the use of prefilled syringe in the study clinic may be eligible to transition from vial and syringe to prefilled syringe dosing. Additionally, regular refresher training on use of prefilled syringe will be provided in study clinic every 24 weeks, and more often as needed.

Subjects should convert their vial and syringe dose to prefilled syringe dose using the following table:

Table 9.4.2.1.2: Conversion from Vial and Syringe Dose to Prefilled Syringe Dose

| Daily Dose (mg)<br>Range | Daily Dose (mg)<br>Round To <sup>a</sup> | # of 2.5mg<br>Prefilled<br>Syringe Needed | # of 10mg<br>Prefilled<br>Syringe Needed | # of 20mg<br>Prefilled<br>Syringe Needed |
|---|---|---|---|---|
| 0 - 3.7 | 2.5 | 1 | 0 | 0 |
| 3.8 - 6.2 | 5 | 2 | | |
| 6.3 - 8.7 | 7.5 | 3 | | |
| 8.8 – 11.2 | 10 | | 1 | |
| 11.3 – 13.7 | 12.5 | 1 | 1 | |
| 13.8 - 16.2 | 15 | 2 | 1 | |
| 16.3 – 18.7 | 17.5 | 3 | 1 | |
| 18.8 - 21.2 | 20 | | | 1 |
| 21.3 - 23.7 | 22.5 | 1 | | 1 |
| 23.8 - 26.2 | 25 | 2 | | 1 |
| 26.3 - 28.7 | 27.5 | 3 | | 1 |
| 28.8 – 31.2 | 30 | | 1 | 1 |
| 31.3 – 33.7 | 32.5 | 1 | 1 | 1 |
| 33.8 – 36.2 | 35 | 2 | 1 | 1 |
| 36.3 – 38.7 | 37.5 | 3 | 1 | 1 |
| 38.8 – 41.2 | 40 | | | 2 |
| 41.3 – 44.9 | 42.5 | 1 | | 2 |
| 45 – 54.9 | 50 | | 1 | 2 |
| 55 – 64.9 | 60 | | | 3 |
| 65 - 74.9 | 70 | | 1 | 3 |
| 75 – 84.9 | 80 | | | 4 |
| 85 – 94.9 | 90 | | 1 | 4 |
| 95 – 104.9 | 100 | | | 5 |
| 105 – 114.9 | 110 | | 1 | 5 |
| 115 – 124.9 | 120 | | | 6 |
| 125 – 134.9 | 130 | | 1 | 6 |
| 135 – 144.9 | 140 | | | 7 |
| 145 – 154.9 | 150 | | 1 | 7 |

<sup>&</sup>lt;sup>a</sup> For <45 mg/day, round to nearest 2.5 mg; for ≥45 mg/day, round to nearest 10 mg.



The excipients in this drug product are tromethamine, tromethamine-hydrochloride, sodium chloride, L-phenylalanine, and water for injection.

rAvPAL PEG doses will be administered SC by either health care professionals or via self-administration. The dose level may be increased or decreased per Investigator determination based on available information regarding a subject's blood Phe level (60 600  $\mu$ mol/L), as well as any adverse events (any hypersensitivity AE) for an individual subject. The dosage that provides control of blood Phe concentrations within the target range of 60-600  $\mu$ mol/L for a minimum of 2 consecutive measurements will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses.

For vial and syringe, drug product packaging will be identified with the lot number and expiration date and will be provided in a box labeled with the study number.

For prefilled syringe, drug product packaging will be identified with the size (2.5 mg, 10 mg, or 20 mg), lot number, and kit identification (ID). The expiration date will be available in a separate Certificate of Compliance issued for each lot.

# 9.4.3 Storage

IP must be stored at  $5 \pm 3$  °C ( $41 \pm 5$  °F) under the conditions specified in the IB. At the site, the IP will be stored in a secure area accessible only to the designated pharmacists and clinical site personnel. All IP must be stored and inventoried and the inventories must be carefully and accurately documented according to applicable state, federal and local regulations, ICH GCP, and study procedures.

Specific instructions for storage of study drug for subjects who qualify for self-administration are provided in the Subject Self-Administration Training Materials.

#### 9.4.4 Directions for Administration

Doses will be administered SC and the favorable dose will be determined for each subject by adjusting the dose level, dose frequency, or both, per the PI, based upon the subject's response to doses. Dosing is up to a maximum dose per week of 5.0 mg/kg (or 375 mg for subjects receiving a fixed dose).

For subjects receiving weight-based dosing, dosage is calculated by multiplying each subject's weight in kilograms (kg) on Day 1 (predose) by the assigned dose (in mg/kg). During the study, if the weight of a subject changes more than 10% from the measurement obtained at baseline or at a previous measurement, the subject's dose may be adjusted to



accommodate the change. The change must be recorded. Refer to the Pharmacy Manual for additional information on calculating dosage.

Subjects who have demonstrated efficacy (as measured by blood Phe within the target range of  $60\text{-}600 \,\mu\text{mol/L}$  for at least 2 consecutive measurements) and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive measurements may be eligible to transition from weight-based dosing to a fixed dosing regimen that would permit daily dosing (5- or 7-days-per-week). Subjects who convert to a fixed-dosing regimen should convert their dose based upon the information presented in Table 9.4.4.1.

Table 9.4.4.1: Fixed Doses for Subjects on Weight-Based Dose Regimen

| Weight-based dose<br>(mg/kg) | Equivalent fixed dose (mg) | Vol for 15 mg/ml concentration (ml) (vial) <sup>a</sup> |
|---|---|---|
| 0.03 | 2.5 | 0.17 |
| 0.06 | 5 | 0.33 |
| 0.12 | 10 | 0.67 |
| 0.25 | 20 | 1.33 |
| 0.5 | 40 | 2.67 |
| 1.0 | 75 | 5 |
| 2.0 | 150 | 10 |
| 3.0 | 225 | 15 |
| 4.0 | 300 | 20 |
| 5.0 | 375 | 25 |

<sup>&</sup>lt;sup>a</sup> Applies to both 1.0 and 1.3 ml withdrawal.

It is preferable that the injection sites should be alternated between doses, ie, upper left arm in Week 1, upper right arm in Week 2, etc. Doses may be administered in any of the common SC areas (upper arm, thigh, abdomen). If dose volume is such that a dose will be divided and given in more than 1 injection site, it is preferable to use both arms, both legs, or both sides of the abdomen.

Subjects may require more than 1 injection per dose, depending upon site policy (ie, some institutions do not permit a single SC injection of greater than 2 mL). Dosage calculations must be performed according to study drug preparation instructions provided in the PAL-003 Pharmacy Manual. Study drug will be administered by clinic staff, other qualified and trained study personnel, or qualified subjects.



Information for dosing of subjects who enroll into this study after completing previous rAvPAL studies is provided in Section 9.1. Instructions for subjects who re-start rAvPAL-PEG dosing due to unplanned missed doses are provided in Section 9.4.10.

Instructions for administration of study drug for subjects who qualify for self-administration are provided in the Subject Self-Administration Training Materials.

## 9.4.5 Method of Assigning Subjects to Treatment Groups

This will be an open-label study; no randomization schedule will be generated.

Subjects will retain the same subject number used in their previous rAvPAL-PEG study.

## 9.4.6 Selection of Doses Used in the Study

This Phase 2 study aims to evaluate the efficacy, safety, tolerability, and PK parameters of multiple doses of rAvPAL-PEG after long-term administration in subjects with PKU. A dose that produces a reduction in blood Phe concentrations to 60-600 µmol/L will be determined for each subject based on preliminary safety, antibody, and efficacy data from this ongoing study.

# 9.4.6.1 Selection of Timing of Dose for Each Subject

Study drug will be administered by clinic staff or other qualified and trained study personnel.

Subjects may self-administer study drug at home if approved by the sponsor's medical monitor and if adequate training is provided (refer to Section 9.4).

## 9.4.7 Blinding

This is an open-label study.

#### 9.4.8 Prior and Concomitant Medications

All prescription and over-the-counter (OTC) medications taken by a subject for 30 days before Screening will be recorded on the designated CRF. The Investigator may prescribe additional medications during the study, as long as the prescribed medication is not prohibited by the protocol. In the event of an emergency, any needed medications may be prescribed without prior approval, but the sponsor's medical monitor must be notified of the use of any contraindicated medications immediately thereafter. Any concomitant medications added or discontinued during the study should be recorded on the CRF.

Use of any investigational product (with the exception of rAvPAL-PEG used in a previous rAvPAL-PEG study) or investigational medical device within 30 days before Screening, or



requirement for any investigational agent prior to completion of all scheduled study assessments, is prohibited.

Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, is prohibited within 6 months prior to Screening and during study participation. A list of PEG-containing injectable drugs is provided in the study reference materials. Subjects who have had a prior hypersensitivity AE to rAvPAL-PEG or a PEG-containing product will be encouraged to be premedicate as outlined in Section 9.1.1. If the hypersensitivity AE worsens with a repeat injection (as determined by the Investigator in consultation with the sponsor's medical monitor) even with premedication prior to study drug dosing, the subject must be withdrawn from the study and complete an Early Termination Visit.

Subjects who have had a prior hypersensitivity AE to rAvPAL-PEG or a PEG-containing product may participate in this study (refer to Section 9.3.2).

Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug is prohibited.

# 9.4.9 Treatment Compliance

The date, time, volume, and concentration of each dose of study drug administered to each subject must be recorded in the dispensing log provided for the study, as well as on the appropriate CRF. This data will be used to assess treatment compliance.

#### 9.4.10 Dose Interruption and Missed Doses

Information for dosing of subjects who enroll into this study after completing previous rAvPAL-PEG studies is provided in Section 9.1.

During this long-term extension study, interruption of rAvPAL-PEG dosing may occur per subject decision or per the Investigator. After a dosing interruption of ≥ four consecutive doses, rAvPAL-PEG administration should be re-started at the same dose level and dosing frequency that was administered prior to the dosing interruption. The first week of dosing of rAvPAL-PEG following a dose interruption should be administered in a clinic setting, and the subject must be observed for 30 minutes following administration due to restarting dosing. Premedication with H1 antagonist, H2 antagonist, and antipyretics (eg, acetaminophen) approximately 2-3 hours prior to study drug should be administered following any dose interruption of ≥ four consecutive doses. If NSAIDs are administered as a premedication, they should be given with food. A follow-up telephone call will be made to the subject to monitor subject safety 24 hours following the return to dosing. Subjects should



continue to perform the study assessments as outlined in the Schedule of Events (refer to Table 9.1.1) during any dosing interruption.

Subjects who miss rAvPAL-PEG dosing due to poor compliance may be discontinued from further study drug per discretion of the Sponsor or Investigator (refer to Section 9.3.3).

# 9.5 Investigational Product Accountability

The PI or designee is responsible for maintaining accurate records (including dates and quantities) of IP received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), IP returned, and IP lost or accidentally or deliberately destroyed. The PI or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

## 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.

Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the PIs study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

Subjects who qualify for self-administration of study drug will be provided with instructions for returning used and unused study drug and the proper disposal of any study drug materials (refer to the Subject Self-Administration Training Materials).

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

# 9.6 Dietary or Other Protocol Restrictions

Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. Subjects who are planning to become pregnant (or impregnate a female partner) may modify their diet in consultation with the investigator and/or study dietician.

Amendment 8: 31 March 2017



A 3-day dietary record will be completed by subjects and will be brought to clinic visits for review with clinic staff. It is preferable that subjects complete the 3-day record immediately prior to their next monthly study visit. The dietary record will be maintained with the study source documents. Information regarding a subject diet diary is provided in Section 9.7.4.

# 9.7 Efficacy and Safety Variables

#### 9.7.1 Efficacy and Safety Measurements Assessed

The Schedules of Events in the Synopsis describe the timing of required evaluations.

For the laboratory assessments, the party responsible for performing the assessment and the pertinent protocol section describing the details of the test are listed in Table 9.7.1.1.

**Section in Protocol for** Party Responsible for **Laboratory Assessment Performing Test Details** Clinical laboratory tests Central laboratory 9.7.6 BioMarin<sup>a</sup> or CRO Antibody testing 9.7.5.2 PK variables BioMarin 9.7.3 Blood Phe concentrations Central laboratory 9.7.2.1 Pregnancy test (urine) and sedimentation Local laboratory 9.7.6. rate 9.7.5.1 9.7.6 Urinalysis Central laboratory

**Table 9.7.1.1: Summary of Laboratory Assessments** 

# 9.7.1.1 Demographic Data and Medical History

Demographic data and a detailed medical history, including allergy history, will be obtained at Screening. The medical history will include specific information concerning any prior or existing medical conditions that might interfere with study participation or safety. This medical history should elicit all major illnesses, diagnoses, and surgeries that the subject has ever had, and whether the subject has a history of alcohol and/or drug abuse.

#### 9.7.1.2 Physical Examination Findings

Physical examination will include assessment of general appearance; CV; dermatologic; head, eyes, ears, nose, and throat; lymphatic; respiratory; GI; musculoskeletal; and neurological/psychological. Other body systems may be examined. Day 1 results will be the baseline values and clinically significant changes from baseline will be recorded as an AE.


Phe, phenylalanine; PK, pharmacokinetic.

<sup>&</sup>lt;sup>a</sup>Analysis of the anti-rAvPAL IgE and anti-rAvPAL-PEG IgE assay will be performed by a Contract Research Organization.



# 9.7.1.3 Vital Sign Measurements

Vital signs will be measured after resting for 5 minutes, and include seated systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in millimeters of mercury (mm Hg), heart rate in beats per minute, respiration rate in breaths per minute, and temperature in degrees Celsius (°C). Height (cm) will be measured at Screening only. Weight will be measured at Screening and then monthly.

## 9.7.1.4 Electrocardiography

A standard 12-lead ECG will be recorded while the subject is resting, at Screening and at the Final Follow-Up (F/U) Visit or Early Termination Visit (ETV). If clinically significant abnormalities are noted at Screening, the PI or designee is required to assess whether it is appropriate for the subject to enroll in the study.

## **9.7.1.5** Chest X-Ray

A chest X-ray will be performed at the Screening, Week 48, and Final Follow-Up (or Early Termination) visits to assess gross pulmonary health.

# 9.7.2 Efficacy Variable

# 9.7.2.1 Blood Phenylalanine Concentrations

Blood samples for Phe concentration measurements will be drawn monthly, at least 2.5 hours after a meal, on the days and time points indicated in the Schedule of Events (Table 9.1.1).

Blood Phe may be collected more often than monthly at the discretion of the Investigator should more frequent monitoring of blood Phe levels be clinically required.

A central laboratory will be used for blood Phe concentration analysis.

#### 9.7.3 Pharmacokinetic Variables

Subjects enrolled in the Substudy will have additional PK sampling performed. For subjects participating in the Substudy, PK sampling will be performed as follows:

- For subjects who are administered rAvPAL-PEG once per week, plasma PK sampling will be performed pre-dose and every 24 hours thereafter (24, 48, 72, and 96 hours if possible), and then pre-dose of the next weekly dose.
- For subjects who are administered rAvPAL-PEG two or three times per week, plasma PK sampling will be performed pre-dose and every 24 hours during the longest period between doses, when possible, and then pre-dose of the next dose.



• For subjects who are administered rAvPAL-PEG four to seven times per week, plasma PK sampling will be performed pre-dose and every 12 hours during the longest period between doses, when possible, and then pre-dose of the next dose.

See Table 9.1.2 for additional details.

BioMarin will perform the analysis.

## 9.7.4 Exploratory Efficacy Variable

Diet will be assessed for its role in blood Phe reduction relative to rAvPAL-PEG dosing using a 3-day diet diary, which will be given to subjects to complete at home. Subjects will bring the completed diary with them to clinic visits on a monthly basis. Subjects will be instructed to record all food, beverages, special low-protein foods, and medical foods consumed for 3 consecutive days each month. If changes in diet are noted per the information on the diet diary, the subject will be instructed to maintain their diet as reported at the beginning of the study or as otherwise instructed by the Investigator.

#### 9.7.5 Safety Variables

## 9.7.5.1 Pregnancy Testing

Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 9.1.1). Subjects who are confirmed to be pregnant per a serum pregnancy test and are temporarily off study drug are not required to perform the scheduled urine pregnancy tests. Female subjects with a positive serum pregnancy test at Screening do not meet eligibility criteria for enrollment.

Additional pregnancy tests will be performed at any visit in which pregnancy status is in question. Serum pregnancy tests will be performed in the event of a positive or equivocal urine pregnancy test result.

Refer to Section 10.3 for details on the reporting procedures to follow in the event of pregnancy.

# 9.7.5.2 Antibody Testing

Immunogenicity will be assessed by determining immune response and neutralizing activity with the following measurements: anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL IgE, anti-rAvPAL-PEG IgE, and anti-rAvPAL-PEG neutralizing antibodies (refer to Section 9.1.1). Immunogenicity assays will be performed at the time points indicated in the Schedule of Events (Table 9.1.1).



BioMarin will perform all antibody testing, except for IgE antibodies, which will be assessed by a Contract Research Organization.

## 9.7.6 Clinical Laboratory Assessments

Any abnormal test results determined to be clinically significant by the Investigator should be repeated (at the Investigator's discretion) until the cause of the abnormality is determined, the value returns to baseline or to within normal limits, or the Investigator determines that the abnormal value is no longer clinically significant. In the event of elevated urinary protein on a test result, a repeat urinalysis should be performed. This repeat urine sample must be performed in the morning at the first or second morning void to allow for accurate test results and may be performed by a home healthcare nurse. Subjects with a confirmed urine/albumin creatinine ratio of  $\geq 100$  mg/g should be referred to a nephrologist for consultation if results were within normal range at baseline. Subjects who had elevated results at baseline followed by a confirmed subsequent increase of 100-200 mg/g from baseline should also be referred to a nephrologist for consultation.

All abnormal clinical laboratory result pages should be initialed and dated by an Investigator, along with a comment regarding whether or not the abnormal result is clinically significant.

The diagnosis, if known, associated with abnormalities in clinical laboratory tests that are considered clinically significant by the Investigator will be recorded on the AE CRF.


PAL-003 A8


# **Table 9.7.6.1: Clinical Laboratory Tests**

| Blood Chemistry | Hematology | Urine Tests <sup>a</sup> | Other |
|---|---|---|---|
| Albumin | Hemoglobin | Appearance | Pregnancy test, if applicable <sup>a</sup> |
| Alkaline Phosphatase | Hematocrit | Color | |
| ALT (SGPT) | WBC count | pН | Phenylalanine |
| AST (SGOT) | RBC count | Specific gravity | Tyrosine |
| Total bilirubin | Platelet count | Ketones | Sedimentation rate <sup>a</sup> |
| BUN | Differential cell count | Protein | |
| Creatinine | | Glucose | |
| GGT | | Spot urine albumin/creatinine ratio | Additional Unscheduled<br>Hypersensitivity Reaction Visit<br>Tests <sup>b</sup> |
| Total protein | | Nitrite | CH50 |
| Calcium | | Urobilinogen | C <sub>1</sub> , C <sub>3</sub> , C <sub>4</sub> |
| Sodium | | Hemoglobin | Serum tryptase level <sup>b</sup> |
| Potassium | | Bilirubin | CRP |
| Glucose | | | Urine N-methyl histamine |
| | | | Urine albumin/creatinine ratio <sup>c</sup> |
| Uric acid | | | Complement Testing <sup>d</sup> |
| CO <sub>2</sub> | | | C <sub>3</sub> |
| Chloride | | | C <sub>4</sub> |

- ALT, alanine aminotransferase; AST, aspartate aminotransferase; BUN, blood urea nitrogen; C, complement; CH50, total hemolytic complement; CO2, carbon dioxide; CRP, C-reactive protein; GGT, gamma-glutamyltransferase; RBC, red blood cell; SGOT, serum glutamic-oxaloacetic transaminase; SGPT, serum glutamic-pyruvic transaminase; WBC, white blood cell.
- <sup>a</sup> To be performed by central laboratory. If urine pregnancy test is positive or equivocal, serum sample will be taken and assessed by a central laboratory. It is recommended that urine samples are obtained as a first or second morning void. In the event of elevated urinary protein on a test result, a repeat urinalysis should be performed. This repeat urine sample must be performed in the morning at the first or second morning void to allow for accurate test results and may be performed by a home healthcare nurse.
- <sup>b</sup> Perform within 24 hours of event onset.
- ° It is recommended that urine samples are obtained as a first or second morning void. Subjects with a confirmed urine/albumin creatinine ratio of  $\geq 100$  mg/g should be referred to a nephrologist for consultation if results were within normal range at baseline. Subjects who had elevated results at baseline followed by a confirmed subsequent increase of 100-200 mg/g from baseline should also be referred to a nephrologist for consultation.
- <sup>d</sup> Complement C<sub>3</sub> and C<sub>4</sub> to be drawn at the Screening Visit and then every 8 weeks or as needed to resolve abnormal test results.

|----------|------------|---------|
|----------|------------|---------|

# 9.7.7 Exploratory Sample Analyses

Blood and urine samples will be collected to evaluate biochemical, molecular, and cellular aspects of PKU and to develop the assays used for these evaluations. For each portion of the blood and urine samples reserved for protocol-specified analyses, there may be multiple sample aliquots. Once samples have been successfully analyzed during the study, unused sample portions may be used during the study or after the subject's study completion for assay development or other purposes.

All samples collected in this study may be used for exploratory research. In addition, samples collected for other purposes may be used for exploratory research use once the primary use has been completed.



#### 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a subject administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (eg, AEs related to screening procedures, medication washout, or no-treatment run-in).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

The study AE reporting period is as follows: After informed consent but prior to initiation of study drug, only SAEs associated with any protocol-imposed interventions will be reported. After informed consent is obtained and the first administration of study drug, all non-serious AEs and SAEs reporting period begins and continues until 4 weeks following the last administration of study drug or the Study Completion Visit/Early Termination Visit, whichever occurs last (refer to Section 12). The criteria for determining, and the reporting of SAEs is provided in Section 10.2.

For this study, a medical device is defined as the prefilled syringe and all of the component parts. The reporting period for device-related events begins with the first dose administered using prefilled syringe and ends with the last dose administered using prefilled syringe. Events assessed by the investigator as related to the device, including malfunction, injury, or medication error, will be captured into an electronic data capture system. All serious events related to the device will be reported to BioMarin Pharmacovigilance (BPV) within 24 hours using the device-related event report form and entered onto the appropriate eCRF page(s) as required.

|----------|------------|---------|
|----------|------------|---------|

The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study drug or study participation is not the cause of the AE. Outcome of AEs (and resolution dates) should be documented on the appropriate CRF page(s) and in the subject's medical record unless the subject is lost to follow-up or it has been determined that the study drug or study participation is not the cause of the AE.

The Investigator responsible for the care of the subject or qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to seriousness, which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

The Investigator will determine the severity of each AE using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.

| Grade | Description |
|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-<br>appropriate instrumental activities of daily living (ADL) <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life-threatening: hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL) <sup>b</sup> |
| 4 | Life threatening or debilitating: consequences; urgent intervention indicated |
| 5 | Death related to AE |

Grade 4 and 5 AEs should always be reported as SAEs.

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

<sup>&</sup>lt;sup>b</sup> Self care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.

| <b>B</b> OMARIN | PAL-003 A8 | Page 72 |
|-----------------|------------|---------|
|-----------------|------------|---------|

The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF, using the categories defined below.

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred OR The administration of the IP and the occurrence of the AE are not reasonably related in time |
| | OR The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts [evidence] or arguments to suggest a causal relationship to the IP. |
| Possibly Related | The administration of the IP and the occurrence of the AE are reasonably related in time AND The AE could be explained equally well by factors or causes other than exposure to the IP. |
| Probably Related | The administration of IP and the occurrence of the AE are reasonably related in time AND The AE is more likely explained by exposure to the IP than by other factors or causes. |

In order to classify AEs and diseases, preferred terms will be assigned by the sponsor to the original terms entered on the CRF, using MedDRA (Medical Dictionary for Regulatory Activities terminology).

Factors suggestive of a causal relationship could include (but are not limited to) the following:

- Plausible temporal relationship
- Absence of alternative explanations
- Rarity of event in a given patient or disease state
- Absence of event prior to study drug exposure
- Consistency with study product pharmacology
- Known relationship to underlying mechanism of study drug action
- Similarity to adverse reactions seen with related drug products
- Abatement of AE with discontinuation of study drug, and/or recurrence of AE with reintroduction of study drug



#### 10.2 Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Is fatal.
- Is life threatening.
  - O Note: Life-threatening refers to an event that places the subject at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Requires or prolongs inpatient hospitalization.
- Results in persistent or significant disability or incapacity.
- Is a congenital anomaly or birth defect in the child or fetus of a subject exposed to IP prior to conception or during pregnancy.
- Important medical events or reactions that may not be immediately life-threatening or
  result in death or hospitalization but may jeopardize the subject or may require
  intervention to prevent one of the other outcomes above should also usually be
  considered serious.

For this protocol, anaphylaxis per NIAID/FAAN criteria for the clinical diagnosis of anaphylaxis is designated as an AE of special interest (serious or nonserious and irrespective of severity) to facilitate rapid reporting and sponsor review. All occurrences of anaphylaxis per NIAID/FAAN criteria will be reported to the sponsor within 24 hours of the site becoming aware of the event using the SAE form. Severity and serious criteria (if applicable) should be reported on the SAE form.

The reporting period for SAEs related to protocol imposed interventions begins after informed consent is obtained, the reporting period for all SAEs begins after first dose of study drug and continues until 4 weeks following the last administration of study drug or End of Treatment Visit. The reporting period for Serious Device Related Events begins after first dose of study drug and ends with the last administered dose.

All SAEs (including serious device-related events), whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event by faxing the study-specific SAE Report Form or device Report Form to BioMarin Pharmacovigilance (BPV). Each SAE must also be reported in the CRF Investigators should not wait to collect information that fully documents the event before notifying BPV of a SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators



submit any information requested by BioMarin as soon as it becomes available. The Investigator should follow all unresolved SAEs until the events are resolved or stabilized, the subject is lost to follow-up, or it has been determined that the study drug or participation is not the cause of the AE. Resolution of AEs (with dates) should be documented in the CRF and in the subject's medical record.

For some SAEs, the Sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).

Reporting of SAEs to the IRB will be done in compliance with the standard operating procedures and policies of the IRB and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB was properly and promptly notified as required.

# 10.3 Adverse Events Occurring Secondary to Other Events

In general, AEs occurring secondary to other events (eg, cascade events) should be identified by their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF. However, medically important events that may be linked and/or separated in time should be recorded as independent events on the eCRF. For example, if severe hemorrhage leads to renal failure, both events should be recorded separately on the eCRF.

#### 10.4 Persistent or Recurrent Adverse Events

A persistent AE is one that extends continuously, without resolution, between subject evaluation time points. Such an event should be recorded only once on the eCRF unless its severity increases or decreases (in which case it should be recorded again on the AE eCRF).

A recurrent AE is one that occurs and resolves between subject evaluation time points, but then subsequently recurs. All recurrences of the AE should be individually recorded as a separate event on the AE eCRF.

### 10.5 Abnormal Laboratory Values

Laboratory test results will be recorded on the laboratory results pages of the eCRF, or appear on electronically produced laboratory reports submitted directly from the central laboratory, if applicable.

Any laboratory result abnormality fulfilling the criteria for a SAE should be reported as such, in addition to being recorded as an AE in the eCRF.

|----------|------------|---------|
|----------|------------|---------|

A clinical laboratory abnormality should be documented as AE if it is not otherwise refuted by a repeat test to confirm the abnormality and any one or more of the following conditions is met:

- Accompanied by clinical symptoms
- Leading to a change in study medication (e.g. dose modification, interruption or permanent discontinuation)
- Requiring a change in concomitant therapy (e.g. addition of, interruption of, discontinuation of, or any other change in a concomitant medication, therapy or treatment).
- The abnormality suggests a disease and/or organ toxicity
- The abnormality is of a degree that requires active management (eg, change of dose, discontinuation of study drug, more frequent follow-up assessments, further diagnostic investigation, etc.)

This applies to any protocol and non-protocol specified safety and efficacy laboratory result from tests performed after the first dose of study medication that falls outside the laboratory reference range and meets the clinical significance criteria.

This does not apply to any abnormal laboratory result that falls outside the laboratory reference range but that does not meet the clinical significance criteria (these will be analyzed and reported as laboratory abnormalities), those that are considered AEs of the type explicitly exempted by the protocol, or those which are a result of an AE that has already been reported.

#### 10.6 Pre-existing Conditions

A pre-existing condition is one that is present at the start of the study. Such conditions should be recorded as medical history on the appropriate eCRF.

A pre-existing condition should be recorded as an AE or SAE during the study only if the frequency, intensity, or character of the condition worsens during the study period. It is important to convey the concept that a pre-existing condition has changed by including applicable language in the verbatim description of the event (eg, more frequent headaches).

# 10.7 General Physical Examination Findings

At screening, any clinically significant abnormality should be recorded as a pre-existing condition (refer to Section 10.6). During the study, any new clinically significant findings and/or abnormalities discovered on physical examination that meet the definition of an AE (or an SAE) must be recorded and document as an AE or SAE on the AE eCRF.



## 10.8 Hospitalization, Prolonged Hospitalization, or Surgery

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as an SAE unless specifically instructed otherwise in this protocol (refer to Section 10.2).

There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include planned hospitalizations or prolonged hospitalizations to the following:

- Perform a protocol-mandated efficacy measurement
- Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed in severity
- Receive scheduled therapy (study drug or otherwise) for the study indication

#### 10.9 Deaths

All deaths that occur during the AE reporting period (refer to Section 10.1 for nonserious AEs and Section 10.2 for SAEs), regardless of attribution, will be recorded on the AE eCRF and expeditiously reported to the Sponsor as an SAE.

When recording a death, the event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the eCRF. If the cause of death is unknown and cannot be ascertained at the time of reporting, record "Unexplained Death" or "Death of Unknown Cause" on the eCRF.

### 10.10 Pregnancy

Pregnancy in a subject or partner should be reported within 24 hours of the site becoming aware of the pregnancy to BioMarin Pharmacovigilance by fax using the Pregnancy Form in the study reference materials. The reporting period for pregnancies begins with informed consent and continues until 4 weeks following the last study drug dose. In addition, pregnancy in a subject is also reported on the Subject Disposition eCRF and the End of Study eCRF if the subject withdraws from the study due to pregnancy. The Investigator must make every effort to follow the subject through resolution of the pregnancy (delivery or termination) and to report the resolution to BPV in the study reference materials. In the event of pregnancy in the partner of a study subject, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.



Abortion, whether therapeutic or spontaneous, should always be classified as an SAE (as the Sponsor considers these to be medically significant), recorded on the eCRF, and expeditiously reported to the Sponsor as an SAE.

# 10.11 Follow-up of Subjects after Adverse Events

For some SAEs and AESIs, the sponsor may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details (eg, hospital discharge summary, consultant report, or autopsy report) deemed necessary to appropriately evaluate the SAE report.

# 10.12 Post-Study Adverse Events

At the last scheduled visit, the investigator should instruct each subject to report to the investigator and/or to BPV directly any subsequent SAEs that the subject's personal physician(s) believes might be related to prior study treatment.

The investigator should notify the study sponsor of any death or SAE occurring at any time after a subject has discontinued or terminated study participation if the investigator believes that the death or SAE may have been related to prior study treatment. The sponsor should also be notified if the investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject who participated in this study.

#### **10.13** Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "...in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV. Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin with 24 hours.

|----------|------------|---------|
|----------|------------|---------|

Examples of situations that may require urgent safety measures include discovery of the following:

- Immediate need to revise the IP administration (i.e., modified dose amount or frequency not defined in protocol).
- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.

# 10.14 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The Investigator is encouraged to discuss with the Sponsor's Medical Office sponsor's medical monitor r any AEs for which the issue of seriousness is unclear or questioned. Contact information for the sponsor's medical monitor is as follows:

Name: MS

Address: 105 Digital Drive

Novato, CA 94949 USA

Phone:

Fax:

E-mail:



#### 11 APPROPRIATENESS OF MEASUREMENTS

# 11.1 Safety and Pharmacokinetics

The PK and safety assessments in this study are used widely and are generally recognized as reliable, accurate, and relevant.

# 11.2 Diet Diary

A 3-day diet diary will be issued to subjects for completion and will be brought to clinic on a monthly basis for review with the clinical study staff. Additional information regarding the diet diary is provided in Section 7.3, and information regarding administration of the diary is provided in Section 9.7.4. Additional information about diet is provided in Section 9.1 and Section 9.6.



#### 12 STUDY PROCEDURES

# 12.1 Prestudy

An ICF must be signed and dated by the subject (or the subject's legally authorized representative if the subject is less than 18 years of age), the PI or designee and witness (if required) before any study-related procedures are performed.

# 12.2 Screening Visit

After subjects have signed an ICF, they will be screened for enrollment into the study. The following study activities will be performed at Screening:

- Medical history, including allergy history, and demographics
- Physical examination
- Vital signs, including height and weight
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Chest X-ray
- 12-lead ECG
- Clinical laboratory tests (including spot urine albumin/creatinine ratio, hematology, chemistry, and urinalysis)
- Complement C<sub>3</sub> and C<sub>4</sub>
- Assessment of SAEs
- Concomitant medications
- Diet query
- Blood Phe and plasma tyrosine concentration

For subjects who participated in a previous rAvPAL-PEG study, these assessments may be the same as those used for the last visit of the previous study, if they occur within 28 days from Day 1.

#### 12.3 Treatment Period

During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications



assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. If there is a skin reaction that lasts  $\geq$  14 days, the Skin Reaction eCRF should be completed and the subject should be referred to a dermatologist for consultation and a skin biopsy. It is recommended that a photograph of the skin reaction may be taken by the subject or the site to help assess the event; photographs may be collected by the sponsor.

If the dose is modified by increasing dose level, additional blood Phe concentration testing should be done daily for 3 days following dose adjustment. If dose is modified by increasing either dose frequency or dose level, additional blood Phe concentration testing should be done prior to each dose for the first 2 weeks following dose adjustment.

# 12.3.1 Day 1 (Week 1)

Within 28 days of completing screening assessments, the following study activities will be performed on Day 1:

- Physical examination
- Vital signs
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.)
- Assessment of SAEs (predose and postdose) and all AEs (postdose)
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- Administer study drug (study drug may be administered on additional days during the week as determined by the Investigator)

## 12.3.2 Weekly Telephone Visit

Subjects should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled visits every 8 weeks per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit:

• Injection-site self inspection (previous and current injection site)

|----------|------------|---------|
|----------|------------|---------|

- Assessment of AEs
- Concomitant medications
- Confirmation of dose level, frequency, and study drug administration

### 12.3.3 Substudy Visits

For subjects participating in the PK substudy, refer to Section 9.7.3 and Table 9.1.2.

# 12.3.4 Every 8 Weeks

Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit.

Visits must be performed in the clinic every 8 weeks. The following study activities will be performed:

- Physical examination
- Vital signs
- Sedimentation rate
- Weight
- Clinical laboratory tests
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.) For safety reasons, this test must be performed prior to the chest X-ray.
- Chest x-ray (Week 48 visit only)
- Complement C<sub>3</sub> and C<sub>4</sub>
- Assessment of AEs
- Concomitant medications
- Diet query
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies)
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the next monthly visit.)

|----------|------------|---------|
|----------|------------|---------|

- Prefilled syringe self-administration training (to be performed prior to subjects transitioning from vial and syringe drug product to prefilled syringe drug product).
- Administer study drug
- Prefilled syringe refresher training (every 24 weeks only)
- If additional training is needed on days subsequent to the 8-week scheduled visit, additional clinic visit(s) or HHRN may be used.

# 12.3.5 Unscheduled Hypersensitivity Reaction Visit

Subjects who have an NCI-CTCAE grade  $\geq 3$  hypersensitivity reaction after rAvPAL-PEG administration (refer to Section 9.1.1) will have assessments performed immediately following (within 24 hours) the reaction.

- Vital signs
- Clinical laboratory tests
- Urine/albumin creatinine ratio
- CRP, CH50, C1, C3, and C4
- Urine N-methyl histamine
- Serum anti-rAvPAL IgE and anti-rAvPAL-PEG IgE only (performed > 8 hours after event onset)
- Serum tryptase level
- Skin biopsy (optional; affected and not affected area; to be performed within 1 week of the reaction)
- Assessment of AEs
- Concomitant medications

Following completion of the Unscheduled Hypersensitivity Reaction visit, subjects may resume study drug administration per the discretion of the Principal Investigator and the sponsor's medical monitor.

# 12.4 Study Completion/Early Termination Visit

Subjects should perform the Study Completion Visit 4 weeks after the last dose of study drug or after completion of study participation, whichever occurs last.

For subjects who terminate from the study early (refer to Section 9.3.3), the Early Termination Visit (ETV) will occur 4 weeks after the final dose of study drug or after

|----------|------------|---------|
|----------|------------|---------|

withdrawal from study participation, whichever occurs last. Subjects who terminate from study drug early should continue to perform the remaining visit assessments in Section 12.3 as applicable until study completion.

Any AE that caused a subject to withdraw from the study or any clinically significant abnormal laboratory value or vital sign measurement identified at the ETV will be followed by the Investigator.

Every reasonable effort should be made to contact any subject who is lost to follow-up.

The following study activities will be performed at the ETV:

- Physical examination
- Vital signs
- 12-lead ECG
- Clinical laboratory tests
- Chest x-ray
- Sedimentation rate
- Urine pregnancy test, if applicable (A serum pregnancy test will be performed in the event of any positive or equivocal urine pregnancy test result.). For safety reasons, this test must be performed prior to the chest X-ray.
- Assessment of AEs
- Concomitant medications
- Diet query
- 3-day diet diary (It is preferable that the subject complete the diary 3 days immediately prior to the Early Termination Visit.)
- PK sample
- Blood Phe and plasma tyrosine concentration
- Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, anti-rAvPAL-PEG neutralizing antibodies)



## 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, CRFs, monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on CRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer CRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 14.1 Statistical and Analytical Plans

Because of the small sample size, no formal statistical tests will be performed. Categorical data will be summarized using frequency and percent, while continuous data will be summarized using descriptive statistics (ie, number of observations, mean, median, standard deviation [SD], minimum, and maximum).

The statistical analysis plan (SAP) will provide additional details about the planned statistical analysis.

# 14.2 Safety Analysis

All subjects who receive any amount of study drug in this study and have postdose safety information will be included in the safety analyses.

The Medical Dictionary for Regulatory Activities terminology (MedDRA) will be used by the sponsor to assign system organ class and preferred term classification to events and diseases based on the original terms entered on the Case Report Form (CRF).

The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity. A by–subject listing will be provided for those subjects who experience a serious AE (SAE), including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose level reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-treatment visits. Changes from baseline to the post-treatment visits will also be provided. Descriptive statistics of vital signs, physical examination results, ECG results, and X-ray results, and immunogenicity test results will also be provided. Additionally, antibodies and titers will be summarized by scheduled time point.

#### 14.3 Pharmacokinetic Analysis

Subjects who complete the Substudy will have the following PK parameters assessed: area under the plasma concentration-time curve (AUC), time to maximum plasma concentration ( $T_{max}$ ), maximum plasma concentration ( $C_{max}$ ), half life ( $t_{1/2}$ ), and clearance (CL/F). Should



data become available from previous rAvPAL-PEG studies that indicate study drug accumulation should also be measured, additional blood draws may be added for PK analysis as needed per the discretion of the Investigator in consultation with the sponsor's medical monitor.

# 14.3.1 Pharmacokinetic Substudy Analysis

For subjects who completed the Substudy, the steady-state PK of rAvPAL-PEG in subjects who have achieved and maintained target blood Phe will be explored. This substudy has been completed as of 20 December 2013.

## 14.4 Efficacy Analysis

Data from all subjects who receive any amount of study drug and who have any post-treatment efficacy data will be included in the efficacy analysis.

Blood Phe concentration at each scheduled time point will be summarized using descriptive statistics (mean, SD, median, minimum, and maximum). Change in blood Phe concentration from baseline (to be defined in the SAP) to each scheduled time point and presence/absence of antibodies will also be summarized. In addition, the proportion of subjects who have maintained target Phe concentrations of  $60\text{-}600~\mu\text{mol/L}$  will be summarized by each scheduled time point.

The relationship of dietary Phe intake (per information reported on the subject diet diary) and blood Phe concentration will also be explored. Subjects who received any amount of study drug with any post-treatment blood Phe concentration measurements and diet diary information will be included in this exploratory analysis.

Details regarding exploratory analyses will be provided in the Statistical Analysis Plan.

#### 14.5 Determination of Sample Size

Subjects who participated in previous rAvPAL-PEG studies may be enrolled into this study. No formal sample size calculation was conducted for this study or the PAL-003 Substudy.

#### 14.6 Handling of Missing Data

All analyses will be presented based on observed data only. Missing data will not be imputed for analyses unless sensitivity analyses are warranted. If imputations are used, detailed imputation methods will be described in the SAP before locking the database.



#### 14.7 Interim Analyses

Safety will be assessed throughout the study on an ongoing basis (refer to Section 15 for information regarding the DMC).

# 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the PI will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an Investigator considers that a subject's safety is compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB must be sought, and the Investigator should inform BioMarin and the full IRB within 2 working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol, and the final SAP, a protocol amendment will not be issued and the SAP will prevail.



## 15 DATA MONITORING COMMITTEE (DMC)

The DMC will act independently in an advisory capacity to BioMarin to monitor the safety of rAvPAL-PEG in subjects who participate in the study.

The responsibilities of the DMC are to:

- Review the study protocol, informed consent and assent documents, and plans for data monitoring.
- Evaluate the progress of the trial, subjects' risk versus benefit, and other factors that could affect the study outcome.
- Assess the effect and relevance of new external evidence.
- Consider relevant information that may have an impact on the safety of the participants or the ethics of the study.
- Protect the safety of the study participants in accordance with the stopping criteria as defined in study protocol Section 9.1.2.
- Make recommendations to the BioMarin concerning continuation or termination of the study or other study modifications based on observations.

|----------|------------|---------|
|----------|------------|---------|

#### 16 COMPENSATION, INSURANCE, AND INDEMNITY

There will be no charge to study subjects to be in this study. BioMarin will pay all costs of tests, procedures, and treatments that are part of this study. In addition, after IRB approval, BioMarin may reimburse the cost of travel for study-related visits. BioMarin will not pay for any hospitalizations, tests, or treatments for medical problems of any sort, whether or not related to the study subject's disease, that are not part of this study. Costs associated with hospitalizations, tests, and treatments should be billed and collected in the way that such costs are usually billed and collected.

The Investigator should contact BioMarin immediately upon notification that a study subject has been injured by the IP or by procedures performed as part of the study. Any subject who experiences a study-related injury should be instructed by the Investigator to seek medical treatment at a pre-specified medical institution if possible, or at the closest medical treatment facility if necessary. The subject should be given the name of a person to contact to seek further information about, and assistance with, treatment for study-related injuries.

The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment, unless the executed Clinical Trial Agreement between BioMarin and the institution of the investigator specifies otherwise. If the subject has followed the Investigator's instructions, BioMarin may pay for reasonable and necessary medical services to treat the injuries caused by the IP or study procedures. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply with the law.



#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic case report forms will be provided for each subject. The Investigator must review and electronically sign the completed CRF casebook to verify its accuracy.

CRFs must be completed using a web-based application that has been validated. Study site personnel will be trained on the application and will enter the clinical data from source documentation. Unless explicitly allowed in the CRF instructions, blank data fields are not acceptable.

In the event of an entry error, or if new information becomes available, the site personnel will correct the value by deselecting the erroneous response and then selecting or entering the factual response. In compliance with 21 CFR Part 11, the system will require the site personnel to enter a reason for changing the value. The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin's policy is that study data on the CRFs must be verifiable to the source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The Investigator must therefore agree to allow direct access to all source data. Subjects (or their legally authorized representative) must also allow access to their medical records, and subjects will be informed of this and will confirm their agreement when giving informed consent.

A CRA designated by BioMarin will compare the CRFs with the original source documents at the study site and evaluate them for completeness and accuracy before designating them as "source data verified" (SDV). If an error is discovered at any time or a clarification is needed, the CRA, or designee, will create an electronic query on the associated field. Site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re—query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject's CRF casebook can be locked, all data fields must be SDV and all queries closed. The Data Manager, or designee, will then set the status of the forms, visits, and the entire casebook to locked. The investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. Upon completion of the clinical study report for the entire study, an electronic copy of each site's casebooks will be copied to a compact disk (CD) and sent to each site for retention with other study documents.



#### 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The PI agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The PI and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin's GCP Compliance Department or designees may conduct an audit of a clinical site at any time during or after completion of the study. The PI will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other Regulatory Agencies may also conduct an audit of the study. If informed of such an inspection, the PI should notify BioMarin immediately. The PI will ensure that the auditors have access to the clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The PI must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The PI must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition or custody of the study files. The PI/institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, including paper copies of study records (e.g., subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the U.S. or an ICH region and until (1) there are no pending or contemplated marketing applications in the United States or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the IP. The PI/institution should retain subject identifiers for at least 15 years after the completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution or private practice, but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should the PI/institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the PI/institution as to when these documents no longer need to be retained.



#### 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages the publication of these data in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Trial Agreement between BioMarin and the Investigator/Institution. Consideration for authorship of all publications will be based on compliance with the Uniform Requirements for Manuscripts Submitted to Biomedical Journals ("Uniform Requirements") of the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org/about-icmje/faqs/icmje-recommendations/) and good publication practices (GPP).



#### 21 REFERENCES

Armstrong, JK, Hempel, G, Koling, S, Chan, LS et. al. Antibody against poly(ethylene glycol) adversely affects PEG-asparaginase therapy in acute lymphoblastic leukemia patients. Cancer 110[1], 103-111. 2007

Brown, SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 114[2], 371-376. 2004

Chen, AM, Scott, MD. Current and future applications of immunological attenuation via pegylation of cells and tissue. BioDrugs 15[12], 833-847. 2001

Davis, S, Abuchowski, A, Park, YK, Davis, FF. Alteration of the circulating life and antigenic properties of bovine adenosine deaminase in mice by attachment of polyethylene glycol. Clin Exp Immunol 46[3], 649-652. 1981

Fisch, RO. Comments on diet and compliance in phenylketonuria. Eur J Pediatr 159 Suppl 2, S142-S144. 2000

Gamez, A, Wang, L, Sarkissian, CN, Wendt, D et. al. Structure-based epitope and PEGylation sites mapping of phenylalanine ammonia-lyase for enzyme substitution treatment of phenylketonuria. Mol Genet Metab 91[4], 325-334. 2007

Ganson, NJ, Kelly, SJ, Scarlett, E, Sundy, JS et. al. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther 8[1], R12. 2006

Guttler, F, Azen, C, Guldberg, P, Romstad, A et. al. Impact of the phenylalanine hydroxylase gene on maternal phenylketonuria outcome. Pediatrics 112[6 Pt 2], 1530-1533. 2003

Harris, JM, Chess, RB. Effect of pegylation on pharmaceuticals. Nat Rev Drug Discov 2[3], 214-221. 2003

Huttenlocher, PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr 159 Suppl 2, S102-S106. 2000

Judge, A, McClintock, K, Phelps, JR, Maclachlan, I. Hypersensitivity and loss of disease site targeting caused by antibody responses to PEGylated liposomes. Mol Ther 13[2], 328-337. 2006

Kaufman, S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr 114[5], 895-900. 1989

Koch, R, Hanley, W, Levy, H, Matalon, K et. al. The Maternal Phenylketonuria International Study: 1984-2002. Pediatrics 112[6 Pt 2], 1523-1529. 2003



Lapis. Long-term Correction of PKU in the Pahenu2 Mouse by Mutant and Chemically Modified Forms of Phenylalanine Ammonium Lyase. ASHG 57th Annual Meeting The American Society of Human Genetics) 2007.

Lee, PJ, Lilburn, M, Baudin, J. Maternal phenylketonuria: experiences from the United Kingdom. Pediatrics 112[6 Pt 2], 1553-1556. 2003

Levy, HL. Historical background for the maternal PKU syndrome. Pediatrics 112[6 Pt 2], 1516-1518. 2003

Matalon, R, Surendran, S, Matalon, KM, Tyring, S et. al. Future role of large neutral amino acids in transport of phenylalanine into the brain. Pediatrics 112[6 Pt 2], 1570-1574. 2003

Richter, AW, Akerblom, E. Antibodies against polyethylene glycol produced in animals by immunization with monomethoxy polyethylene glycol modified proteins. Int Arch Allergy Appl Immunol 70[2], 124-131. 1983

Richter, AW, Akerblom, E. Polyethylene glycol reactive antibodies in man: titer distribution in allergic patients treated with monomethoxy polyethylene glycol modified allergens or placebo, and in healthy blood donors. Int Arch Allergy Appl Immunol 74[1], 36-39. 1984

Rouse, B, Azen, C. Effect of high maternal blood phenylalanine on offspring congenital anomalies and developmental outcome at ages 4 and 6 years: the importance of strict dietary control preconception and throughout pregnancy. J Pediatr 144[2], 235-239. 2004

Sampson, HA, Munoz-Furlong, A, Campbell, RL, Adkinson, NF, Jr. et. al. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol 117[2], 391-397. 2006

Scott, MD, Murad, KL, Koumpouras, F, Talbot, M et. al. Chemical camouflage of antigenic determinants: stealth erythrocytes. Proc Natl Acad Sci U S A 94[14], 7566-7571. 1997

Scriver, CR, Kaufman. Hyperphenylalaninemia: Phenylalanine Hydroxylase Deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and Molecular Bases of Inherited Disease. New York: McGraw-Hill, 2001: 1667-1724.

Walter, JH, White, FJ, Hall, SK, MacDonald, A et. al. How practical are recommendations for dietary control in phenylketonuria? Lancet 360[9326], 55-57. 2002

Webster, R, Didier, E, Harris, P, Siegel, N et. al. PEGylated proteins: evaluation of their safety in the absence of definitive metabolism studies. Drug Metab Dispos 35[1], 9-16. 2007



#### 22 INVESTIGATOR RESPONSIBILITIES

## 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and institutional review board (IRB) review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68.
- He or she will ensure that the IRB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB. Additionally, he or she will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.



#### 23 SIGNATURE PAGE

**Protocol Title:** Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects with PKU

Protocol Number: PAL-003, Amendment 8

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me

| Investigator Signature | Date |
|------------------------|------|
| Printed name: | |

# Accepted for the Sponsor:



|----------|------------|---------|--|
|----------|------------|---------|--|

### 24 PROTOCOL AMENDMENT TEXT REVISIONS

The following is a summary of significant protocol revisions; added text is <u>underlined</u> and deleted text is <u>struck</u>. Additional administrative changes have been made for consistency and clarity throughout this amendment and are reflected in the protocol body. Revisions made to the Synopsis (Section 2) are reflected in the corresponding protocol section as appropriate. Revisions to cross references to protocol tables, figures, sections, and references reside within the protocol body.

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Global change | Up to 102 Approximately 119 weeks | 9 |
| Global change | Premedication with H1 antagonist, H2 antagonist, and non-steroidal anti-inflammatory medication (NSAIDs)antipyretics (eg. acetaminophen) approximately 2-3 hours prior to study drug should be administered for 1 week upon reintroduction of study drug at Part 3, Week 1 and Part 4, Week 1, as well as upon reintroduction of study drug after resolution of an AE, following any dose interruption of ≥ 4 days, and for any dose increases in Part 4. If non-steroidal anti-inflammatory medication (NSAIDs) is administered as a premedication, it NSAIDs should be given with food and may be omitted if not tolerated. | 6 |
| Section 7.4.1, Toxicity Due to Exposure to Polyethylene Glycol (PEG) | Based on phase 3 data, as of 4MAR2016, there have been no reported events of glomerulonephritis or renal failure reported with pegvaliase administration. Of the 10 subjects identified with UAC ratios ≥ 3 mg/mmol on 3 or more consecutive measurements, values were generally in the microalbuminuria range and none had concurrent sustained hematuria. Seven of these 10 subjects had microalbuminuria at baseline prior to pegvaliase exposure, of which 2 events resolved while on pegvaliase treatment and 4 events did not progress while subjects remained on pegvaliase. One of these 7 subjects with baseline microalbuminuria (3.62 mg/mmol at baseline) had an increase in their UAC ratio during the study, which was more apparent after dose titration to 60 mg of pegvaliase (remaining in microalbuminuria range, with a most recent value of 20.36 mg/mmol), however evaluating relationship to pegvaliase treatment is confounded | 1 |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | by a medical history of obesity, hypertension, and new onset pre-diabetes during the Phase 3 | |
| | study that are conditions also associated with development of microalbuminuria. The subject | |
| | continues on pegvaliase treatment with continued safety monitoring. | |
| | Three of the 10 subjects developed new onset microalbuminuria for at least 3 consecutive | |
| | measurements during the Phase 3 study, one of which resolved while continuing on pegvaliase | |
| | treatment and 1 subject continues to have fluctuating low level microalbuminuria with intermittent | |
| | values in the normal range. One subject discontinued from the Phase 3 study after a few | |
| | intermittent elevations into the microalbuminuria range. The subject had a maximum UAC ratio of | |
| | 175 mg/g on Day 8 on the study; at the time of study and study drug discontinuation (Day 36), | |
| | UAC ratio was within the normal range at 19 mg/g. The final study visit recorded for this subject | |
| | (Day 67) had a UAC ratio of 17 mg/g. This subject reported a single concurrent grade 1 event of | |
| | urticaria, which resolved in 2 days, and no other reported events suggestive of immune complex | |
| | disease. None of the subjects described above have developed sustained elevations in serum | |
| | creatinine or concurrent sustained hematuria. | |
| | To monitor for renal toxicity, subjects participating in this study will undergo urinalysis, will be | |
| | assessed for urine albumin/creatinine ratio, and will undergo blood chemistry tests to assess renal | |
| | function. In this study, subjects will be monitored closely with urine examinations and blood | |
| | chemistries to follow kidney function. | |
| Section 9.1, Overall Study<br>Design and Plan | A subject will continue in PAL-003 until one of the following occurs: | 9 |
| Design and Flan | • The subject has completed the study through the Month 98 Week 476 visit. | |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Section 9.1, Overall Study | Because the risks of taking BMN 165 during pregnancy and breastfeeding are unknown, subjects | 2 |
| Design and Plan | cannot take BMN 165 if they are trying to conceive, are pregnant, or are breastfeeding. Male | |
| | subjects who are planning to impregnate a female partner and female subjects who are trying to | |
| | become pregnant during the study will be discontinued immediately from study drug. Male | |
| | subjects who have impregnated a female partner may re start study drug after conception but must | |
| | return to the study required contraception use, which must include one barrier method. During | |
| | Part 4 only, subjects who remain in the study after discontinuation of study drug due to pregnancy | |
| | may re introduce BMN 165 dosing after the birth has been reported (or termination of the | |
| | pregnancy) and breastfeeding has completed (if applicable) or after the subject is no longer | |
| | actively trying to conceive. Re starting BMN 165 dosing must be per investigator and sponsor | |
| | agreement based on an assessment of the known risks and potential benefits while taking BMN | |
| | 165. Female subjects must return to the study required contraception use, which must include one | |
| | barrier method, immediately after the birth (or termination of the pregnancy). | |
| | Because the risks of taking BMN 165 during pregnancy and breastfeeding are unknown, subjects cannot take BMN | |
| | 165 if they are trying to conceive, are pregnant, or are breastfeeding (refer to Section 9.3.2 for Exclusion Criteria). | |
| | Male subjects who are planning to impregnate a female partner and female subjects who are trying to become | |
| | pregnant during the study must be temporarily discontinued from study drug for 4 weeks prior to trying to conceive. | |
| | During that time, subjects must use two acceptable methods of contraception. Subjects who are planning to become pregnant (or impregnate a female partner) may modify their diet in consultation with the investigator and/or study | |
| | dietician. Subjects who are confirmed to be pregnant per a serum pregnancy test and are temporarily off study drug | |
| | are not required to perform the scheduled urine pregnancy tests. Subjects who are pregnant or are trying to conceive | |
| | and have temporarily discontinued study drug should not perform the scheduled PK assessments. Male subjects who | |
| | have impregnated a female partner may re-start study drug after conception following the investigator's consultation | |
| | with and approval by the medical monitor. Male subjects must return to the study-required contraception use (refer to | |
| | Section 9.3.1 for Inclusion Criteria), which must include one barrier method, prior to restarting study drug. Female | |
| | subjects who remain in the study after temporary discontinuation of study drug due to pregnancy may restart BMN | |
| | 165 dosing after a confirmed negative urine pregnancy test result, the birth has been reported (or termination of the | |
| | pregnancy), and breastfeeding has completed (if applicable) or after the subject is no longer actively trying to | |
| | conceive. Re-starting BMN 165 dosing requires the investigator's prior consultation with and approval by the medical | |
| | monitor. Female subjects must return to the study-required contraception use (refer to Section 9.3.1), which must | |
| | <u>include one barrier method, immediately after the birth (or termination of the pregnancy).</u> | |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Section 9.1, Table 9.1.1,<br>Schedule of Events | The Schedule of Event tables have been updated to reflect the changes in this amendment. Additionally, the monthly visits have been modified to occur every 8 weeks. | 8, 11 |
| Section 9.1.1, Response to<br>Hypersensitivity Adverse<br>Events | Subjects who experience an injection-site skin reaction that lasts ≥ 14 days should be referred to a dermatologist for consultation and a skin biopsy. | 5 |
| Section 9.6, Dietary or<br>Other Protocol<br>Restrictions | Subjects will be instructed that diet should not be altered during the course of the study. Any decision to modify subject diet must be made per the Investigator and must be performed under the supervision of the Investigator. Subjects who are planning to become pregnant (or impregnate a female partner) may modify their diet in consultation with the investigator and/or study dietician. | 2 |
| Section 9.7.5.1, Pregnancy<br>Testing | Female subjects of childbearing potential will have a urine pregnancy test at the time points specified in the Schedules of Events (Table 9.1.1). Subjects who are confirmed to be pregnant per a serum pregnancy test and are temporarily off study drug are not required to perform the scheduled urine pregnancy tests. | 2 |
| Section 9.7.5.2, Antibody<br>Testing | BioMarin or CRO will perform all antibody testing, except for IgE antibodies, which will be assessed by a Contract Research Organization. | 11 |
| Section 9.7.6, Clinical<br>Laboratory Assessments | Any abnormal test results determined to be clinically significant by the investigator should be repeated (at the discretion of the investigator) until the cause of the abnormality is determined, the value returns to the level from Day 1 of Part 2 or to within normal limits, or the investigator determines that the abnormal value is no longer clinically significant. In the event of elevated urinary protein on a test result, a repeat urinalysis should be performed. This repeat urine sample must performed in the morning at the first or second morning void to allow for accurate test results and may be performed by a home healthcare nurse. Subjects with a confirmed urine/albumin creatinine ratio of $\geq 100$ mg/g should be referred to a nephrologist for consultation | 1, 4 |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | if results were within normal range at baseline. Subjects who had elevated results at baseline | |
| | followed by a confirmed subsequent increase of 100-200 mg/g from baseline should also be | |
| | referred to a nephrologist for consultation. | |
| Section 9.7.6.1, Table 9.7.6.1.1 (Clinical | The table has been revised to add the following footnotes: | 1, 4 |
| Laboratory Tests) | <sup>a</sup> To be performed by central laboratory. If urine pregnancy test is positive or equivocal, serum | |
| | sample will be taken and assessed by a central laboratory. It is recommended that urine samples | |
| | are obtained as a first or second morning void. In the event of elevated urinary protein on a test | |
| | result, a repeat urinalysis should be performed. This repeat urine sample must performed in the | |
| | morning at the first or second morning void to allow for accurate test results and may be | |
| | performed by a home healthcare nurse. | |
| | <sup>c</sup> It is recommended that urine samples are obtained as a first or second morning void. Subjects | |
| | with a confirmed urine/albumin creatinine ratio of ≥ 100 mg/g should be referred to a | |
| | nephrologist for consultation if results were within normal range at baseline. Subjects who had | |
| | elevated results at baseline followed by a confirmed subsequent increase of 100-200 mg/g from | |
| | baseline should also be referred to a nephrologist for consultation. | |
| Section 9.7.7, Exploratory | Blood and urine samples will be collected to evaluate biochemical, molecular, and cellular aspects | 7 |
| Sample Analyses | of PKU and to develop the assays used for these evaluations. For each portion of the blood and | |
| | urine samples reserved for protocol-specified analyses, there may be multiple sample aliquots. | |
| | Once samples have been successfully analyzed during the study, unused sample portions may be | |
| | used during the study or after the subject's study completion for assay development or other | |
| | purposes. | |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | All samples collected in this study may be used for exploratory research. In addition, samples collected for other purposes may be used for exploratory research use once the primary use has been completed. | |
| Section 10.1., Adverse<br>Events | Factors suggestive of a causal relationship could include (but are not limited to) the following: Plausible temporal relationship Absence of alternative explanations Rarity of event in a given patient or disease state Absence of event prior to study drug exposure Consistency with study product pharmacology Known relationship to underlying mechanism of study drug action Similarity to adverse reactions seen with related drug products Abatement of AE with discontinuation of study drug, and/or recurrence of AE with | 3 |
| Section 10.3, Adverse Events Occurring | In general, AEs occurring secondary to other events (eg, cascade events) should be identified by | 3 |
| Secondary to Other<br>Events | their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF. However, medically important events that may be linked and/or separated in time should be recorded as independent events on the eCRF. For example, if severe hemorrhage leads to renal failure, both events should be recorded separately on the eCRF. | |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Section 10.4, Persistent or<br>Recurrent Adverse<br>Events | A persistent AE is one that extends continuously, without resolution, between subject evaluation time points. Such an event should be recorded only once on the eCRF unless its severity increases or decreases (in which case it should be recorded again on the AE eCRF). A recurrent AE is one that occurs and resolves between subject evaluation time points, but then subsequently recurs. All recurrences of the AE should be individually recorded as a separate event on the AE eCRF. | 3 |
| Section 10.5, Abnormal Laboratory Values | Laboratory test results will be recorded on the laboratory results pages of the eCRF, or appear on electronically produced laboratory reports submitted directly from the central laboratory, if applicable. Any laboratory result abnormality fulfilling the criteria for a SAE should be reported as such, in addition to being recorded as an AE in the eCRF. A clinical laboratory abnormality should be documented as AE if it is not otherwise refuted by a repeat test to confirm the abnormality and any one or more of the following conditions is met: • Accompanied by clinical symptoms • Leading to a change in study medication (e.g. dose modification, interruption or permanent discontinuation) • Requiring a change in concomitant therapy (e.g. addition of, interruption of, discontinuation of, or any other change in a concomitant medication, therapy or treatment). • The abnormality suggests a disease and/or organ toxicity | 3 |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | The abnormality is of a degree that requires active management (eg, change of dose, discontinuation of study drug, more frequent follow-up assessments, further diagnostic investigation, etc.) | |
| | This applies to any protocol and non-protocol specified safety and efficacy laboratory result from tests performed after the first dose of study medication that falls outside the laboratory reference range and meets the clinical significance criteria. | |
| | This does not apply to any abnormal laboratory result that falls outside the laboratory reference range but that does not meet the clinical significance criteria (these will be analyzed and reported as laboratory abnormalities), those that are considered AEs of the type explicitly exempted by the protocol, or those which are a result of an AE that has already been reported. | |
| Section 10.6, Pre-existing Conditions | A pre-existing condition is one that is present at the start of the study. Such conditions should be recorded as medical history on the appropriate eCRF. A pre-existing condition should be recorded as an AE or SAE during the study only if the frequency, intensity, or character of the condition worsens during the study period. It is important to convey the concept that a pre-existing condition has changed by including applicable language in the verbatim description of the event (eg, more frequent headaches). | 3 |
| Section 10.7, General<br>Physical Examination<br>Findings | At screening, any clinically significant abnormality should be recorded as a pre-existing condition (refer to Section 10.6). During the study, any new clinically significant findings and/or abnormalities discovered on physical examination that meet the definition of an AE (or an SAE) must be recorded and document as an AE or SAE on the AE eCRF. | 3 |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Section 10.8, Hospitalization, Prolonged Hospitalization, or Surgery | Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as an SAE unless specifically instructed otherwise in this protocol (refer to Section 10.2). There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include planned hospitalizations or prolonged hospitalizations to the following: • Perform a protocol-mandated efficacy measurement • Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed • Receive scheduled therapy (study drug or otherwise) for the study indication | 3 |
| Section 10.9, Deaths | All deaths that occur during the AE reporting period (refer to Section 10.1 for nonserious AEs and Section 10.2 for SAEs), regardless of attribution, will be recorded on the AE eCRF and expeditiously reported to the Sponsor as an SAE. When recording a death, the event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the eCRF. If the cause of death is unknown and cannot be ascertained at the time of reporting, record "Unexplained Death" or "Death of Unknown Cause" on the eCRF. | 3 |
| Section 10.10, Pregnancy | Pregnancy in a subject or partner should be reported to BPV within 24 hours of the site becoming aware of the pregnancy by faxing the Pregnancy Form in the study reference materials. The reporting period for pregnancies begins with informed consent and continues until 4 weeks following the last study drug dose or the End of Treatment visit. In addition, pregnancy in a subject should also be reported on the End of Study eCRF and the Subject Disposition eCRF if the subject withdraws from the study due to pregnancy | 3 |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | Abortion, whether therapeutic or spontaneous, should always be classified as an SAE (as the | |
| | Sponsor considers these to be medically significant), recorded on the eCRF, and expeditiously | |
| | reported to the Sponsor as an SAE. | |
| Section 10.11, Follow-up | For some SAEs and AESIs, the sponsor may follow up by telephone, fax, electronic mail, and/or a | 3 |
| of Subjects after Adverse<br>Events | monitoring visit to obtain additional case details (eg, hospital discharge summary, consultant | |
| Dvents | report, or autopsy report) deemed necessary to appropriately evaluate the SAE report. | |
| Section 10.12, Post-Study | At the last scheduled visit, the investigator should instruct each subject to report to the | 3 |
| Adverse Events | investigator and/or to BPV directly any subsequent SAEs that the subject's personal physician(s) | |
| | believes might be related to prior study treatment. | |
| | The investigator should notify the study sponsor of any death or SAE occurring at any time after a | |
| | subject has discontinued or terminated study participation if the investigator believes that the | |
| | death or SAE may have been related to prior study treatment. The sponsor should also be notified | |
| | if the investigator should become aware of the development of cancer or of a congenital anomaly | |
| | in a subsequently conceived offspring of a subject who participated in this study. | |
| Section 10.14, BioMarin | Name: | 10 |
| Pharmacovigilance<br>Contact Information | Address: 105 Digital Drive | |
| Contact Information | Novato, CA 94949 USA | |
| | Phone: | |
| | Fax: | |
| | E-mail: | |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Section 12.3, Treatment Period | During the Treatment Period, additional visits may occur if deemed necessary to monitor AEs or blood Phe concentrations. On days that a dose is given, assessments will be done predose unless otherwise specified. Subjects must have AEs and concomitant medications assessed whenever dose is administered even if the administration does not coincide with a scheduled clinic visit. If there is a skin reaction that lasts ≥ 14 days, the Skin Reaction eCRF should be completed and the subject should be referred to a dermatologist for consultation and a skin biopsy. It is recommended that aA photograph of the skin reaction may be taken by the subject or the site to help assess the event; photographs and may be collected by the sponsor. | 5 |
| Section 12.3.2, Weekly<br>Telephone Visit | Subjects should have a weekly telephone visit conducted. Subjects must still come into the clinic for the scheduled monthly visits every 8 weeks per Table 9.1.1. The following should be discussed with the subject during the weekly telephone visit: | 8 |
| Section 12.3.4, Every 8<br>Weeks | Beginning with Week 4, monthly vVisits must be performed in the clinic every 8 weeks. The following study activities will be performed: • Physical examination • Sedimentation rate • Complement C <sub>3</sub> and C <sub>4</sub> • PK sample • Serum anti-rAvPAL-PEG antibodies (anti-PAL IgG, anti-PAL IgM, anti-PEG IgG, anti-PEG IgM, and anti-rAvPAL-PEG neutralizing antibodies) • Prefilled syringe refresher training (every 24 weeks only) • If additional training is needed on days subsequent to the monthly 8-week scheduled visit, additional clinic visit(s) or HHRN may be used. | 8 |

|----------|------------|----------|
|----------|------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Section 12.3.5, Quarterly Visits | This section has been deleted. | 8 |
| Section 17, Case Report<br>Forms and Source<br>Documents | Before a CRF casebook can be locked, data fields must be source data verified and queries closed. The investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. The Data Manager (or designee) will then set the status of the forms, visits, and the entire casebook to Locked. The investigator will then electronically sign the casebook, specifying that the information on the CRFs is accurate and complete. Upon completion of the clinical study report, an electronic copy of each site's casebooks will be copied to a compact disk and will be sent to each site for retention with other study documents. | 11 |